Comparative Effectiveness of Tirzepatide and Semaglutide in Patients With Low, Moderate, and High Cardiovascular Risk with Type 2 Diabetes and Obesity

NCT07096063

**10<sup>th</sup> August 2025** 

| Research question & Objectives | Comparative effectiveness of semaglutide and tirzepatide in patients at low, moderate, and high cardiovascular risk with type 2 diabetes and obesity: Tirzepatide vs Semaglutide in Individuals at Cardiovascular Risk This study is part of a three-stage project evaluating the comparative effectiveness of semaglutide and tirzepatide in patients at low, moderate, and high cardiovascular risk with type 2 diabetes and obesity: The aim of this study is to assess the comparative effectiveness of tirzepatide vs dulaglutide, semaglutide vs sitagliptin, and tirzepatide vs semaglutide on the risk of major adverse cardiovascular events (MACE) among individuals typically treated in clinical practice who are at low, moderate, and high cardiovascular risk with type 2 diabetes and overweight. |
|---|---|
| Protocol version | Version 2 |
| Last update date | August 10, 2025 |
| Contributors | Primary investigators contact information: Dr. Nils Krüger, nkruger1@bwh.harvard.edu Dr. Shirley Wang, swang1@bwh.harvard.edu Contributor names: Dr. Krüger implemented the study design in the Aetion Evidence Platform. He is responsible for the validity of the design and analytic choices. All implementation steps are recorded and the implementation history is archived in the platform. |
| Study registration | Site: clinicaltrials.gov<br>Identifier: NCT07096063 |
| Sponsor | Organization: N/A<br>Contact: N/A |

| Conflict of interest | Dr. Krüger has no conflict of interest. |
|----------------------|-------------------------------------------------|
| | Dr. Wang has consulted for Cytel Incs, Exponent |
| | Inc, and MITRE an FFRDC for Centers for |
| | Medicare and Medicaid for unrelated work. |

# **Table of contents**

| A mendments and updates 6. Remain and background 6. Research question and objectives 7. Table 2. Primary and secondary research questions and objectives 7. Table 2. Primary and secondary research questions and objectives 7. Table 2. Primary and secondary research questions and objectives 7. Table 2. Primary and secondary research questions and objectives 7. Table 2. Primary and secondary research questions and objectives 19. Castudy design diagrams for the comparison of tirzepatide vs dulaglutide, semaglutide vs sitagliptin, and tirzepatide vs semaglutide. 20. Castudy design diagrams for the comparison of tirzepatide vs dulaglutide, semaglutide vs sitagliptin, and tirzepatide vs semaglutide. 20. Castudy design diagrams for the comparison of tirzepatide vs dulaglutide, semaglutide vs sitagliptin, and tirzepatide vs semaglutide. 20. Castudy design diagrams for the comparison of tirzepatide vs dulaglutide, semaglutide vs sitagliptin, and tirzepatide vs semaglutide. 20. Castudy design diagrams for the comparison of tirzepatide vs dulaglutide, semaglutide vs sitagliptin, and tirzepatide vs semaglutide. 20. Castudy design diagrams for the comparison of tirzepatide vs dulaglutide, semaglutide vs sitagliptin, and tirzepatide vs semaglutide. 20. Castudy design diagrams for the comparison of tirzepatide vs dulaglutide, semaglutide vs sitagliptin, and tirzepatide vs semaglutide. 20. Castudy design diagrams for the comparison of tirzepatide vs dulaglutide, semaglutide vs sitagliptin, and tirzepatide vs semaglutide. 20. Castudy design diagrams for the comparison of tirzepatide vs dulaglutide, semaglutide vs sitagliptin, and tirzepatide vs semaglutide. 20. Castudy design diagrams for the comparison of tirzepatide vs dulaglutide, semaglutide vs sitagliptin, and tirzepatide vs semaglutide vs sita | I. Title Page | 1 |
|---|---|---|
| Rationale and background Research question and objectives Table 2. Primary and secondary research questions and objectives Research methods 6.1 Study design 6.1 Study design 6.2 Study design idiagrams for the comparison of tirzepatide vs dulaglutide, semaglutide vs sitagliptin, and tirzepatide vs semaglutide vs setting 6.3 Stetting 6.3.1 Context and rationale for definition of time 0 (and other primary time anchors) for entry to the study population 21 6.3.2 Context and rationale for study inclusion criteria: 6.3.3 Context and rationale for study exclusion criteria: 6.3.4 Variables 6.4.4 Variables 6.4.2 Context and rationale for exposure(s) of interest 6.4.2 Context and rationale for outcome(s) of interest 6.4.3 Context and rationale for outcome(s) of interest 6.4.4 Context and rationale for follow-up 7 Table 2. Operational Definitions of follow-up 7 Table 2. Operational Definitions of Covariates (confounding variables and effect modifiers, e.g. risk factors, comorbidities, comedications) 8 Context and rationale for analysis plan 7 Table 3. Primary, secondary, and subgroup analysis specification 7 Table 4. Sensitivity analyses – rationale, strengths and limitations 6.6 Data sources 6.6 Data sources 6.7 Data management 6.8 Quality control 6.9 Study size and feasibility 7 Limitation of the methods | 2. Abstract | 5 |
| Table 2. Primary and secondary research questions and objectives 7 Table 2. Primary and secondary research questions and objectives 7 Seesarch methods 19 6.1 Study design diagrams for the comparison of tirzepatide vs dulaglutide, semaglutide vs sitagliptin, and tirzepatide vs semaglutide. 20 6.3 Setting 21 6.3.1 Context and rationale for definition of time 0 (and other primary time anchors) for entry to the study population 21 6.3.2 Context and rationale for study inclusion criteria: 22 6.3.3 Context and rationale for study exclusion criteria: 22 6.4.4 Variables 22 6.4.4 Context and rationale for exposure(s) of interest 22 6.4.2 Context and rationale for outcome(s) of interest 22 6.4.2 Context and rationale for follow-up 23 7 able 1. Operational Definitions of follow-up 23 6.4.4 Context and rationale for covariates (confounding variables and effect modifiers, e.g. risk factors, comorbidities, comedications) 25 7 able 2. Operational Definitions of Covariates 25 6.5. Data analysis 42 6.5.1 Context and rationale for analysis plan 42 7 able 3. Primary, secondary, and subgroup analysis specification 42 7 able 4. Sensitivity analyses – rationale, strengths and limitations 55 6.6.1 Context and rationale for data sources 55 6.6.1 Context and rationale for data sources 55 6.6.2 Data management 56 6.8 Quality control 58 6.9 Study size and feasibility 59 7. Limitation of the methods 59 | 3. Amendments and updates | 5 |
| Table 2. Primary and secondary research questions and objectives 5. Research methods 6.1 Study design 6.2 Study design diagrams for the comparison of tirzepatide vs dulaglutide, semaglutide vs sitagliptin, and tirzepatide vs semaglutide. 6.3 Setting 7 6.3 Setting 7 6.3.1 Context and rationale for definition of time 0 (and other primary time anchors) for entry to the study population 7 6.3.2 Context and rationale for study exclusion criteria: 6.3.3 Context and rationale for study exclusion criteria: 6.3.4 Context and rationale for exposure(s) of interest 6.4 Variables 6.4.1 Context and rationale for exposure(s) of interest 6.4.2 Context and rationale for outcome(s) of interest 6.4.3 Context and rationale for follow-up 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 | 4. Rationale and background | 6 |
| 6. Research methods 6.1 Study design 6.2 Study design flagrams for the comparison of tirzepatide vs dulaglutide, semaglutide vs sitagliptin, and tirzepatide vs semaglutide. 6.3 Setting 6.3 Setting 6.3.1 Context and rationale for definition of time 0 (and other primary time anchors) for entry to the study population 21 6.3.2 Context and rationale for study inclusion criteria: 6.3.3 Context and rationale for study exclusion criteria 6.3.3 Context and rationale for exposure(s) of interest 6.4.4 Variables 6.4.1 Context and rationale for outcome(s) of interest 6.4.2 Context and rationale for outcome(s) of interest 6.4.3 Context and rationale for follow-up 23 7 able 1. Operational Definitions of follow-up 7 able 2. Operational Definitions of Covariates (confounding variables and effect modifiers, e.g. risk factors, comorbidities, comedications) 7 able 2. Operational Definitions of Covariates 6.5 Data analysis 6.5.1 Context and rationale for analysis plan 42 6.5.2 Context and rationale for analysis plan 42 7 able 3. Primary, secondary, and subgroup analysis specification 42 7 able 4. Sensitivity analyses – rationale, strengths and limitations 6.6 Data sources 6.6.1 Context and rationale for data sources 7 55 7 able 5. Metadata about data sources and software 6.7 Data management 6.8 Quality control 6.8 Quality control 6.9 Study size and feasibility 59 7 Limitation of the methods | 5. Research question and objectives | 7 |
| 6.1 Study design 19 6.2 Study design diagrams for the comparison of tirzepatide vs dulaglutide, semaglutide vs sitagliptin, and tirzepatide vs semaglutide. 20 6.3 Setting 21 6.3.1 Context and rationale for definition of time 0 (and other primary time anchors) for entry to the study population 21 6.3.2 Context and rationale for study inclusion criteria: 22 6.3.3 Context and rationale for study exclusion criteria 22 6.4 Variables 22 6.4.1 Context and rationale for exposure(s) of interest 22 6.4.2 Context and rationale for outcome(s) of interest 22 6.4.3 Context and rationale for follow-up 23 7 able 1. Operational Definitions of follow-up 23 6.4.4 Context and rationale for covariates (confounding variables and effect modifiers, e.g. risk factors, comorbidities, comedications) 25 6.5 Data analysis 42 6.5.1 Context and rationale for analysis plan 42 Table 3. Primary, secondary, and subgroup analysis specification 42 Table 4. Sensitivity analyses – rationale, strengths and limitations 55 6.6 Data sources 55 6.6.1 Context and rationale for data sources 55 7 able 5. Metadata about data sources and software 56 6.7 Data management 56 6.8 Quality control 58 6.9 Study size and feasibility 59 7. Limitation of the methods | Table 2. Primary and secondary research questions and objectives | 7 |
| 6.2 Study design diagrams for the comparison of tirzepatide vs dulaglutide, semaglutide vs sitagliptin, and tirzepatide vs semaglutide. 20 6.3 Setting 21 6.3.1 Context and rationale for definition of time 0 (and other primary time anchors) for entry to the study population 21 6.3.2 Context and rationale for study inclusion criteria: 22 6.3.3 Context and rationale for study exclusion criteria: 22 6.4 Variables 22 6.4.1 Context and rationale for exposure(s) of interest 22 6.4.2 Context and rationale for outcome(s) of interest 22 6.4.3 Context and rationale for outcome(s) of interest 22 6.4.4 Context and rationale for coursels of follow-up 23 6.4.4 Context and rationale for covariates (confounding variables and effect modifiers, e.g. risk factors, comorbidities, comedications) 25 6.5 Data analysis 42 6.5.1 Context and rationale for analysis plan 42 Table 3. Primary, secondary, and subgroup analysis specification 42 Table 4. Sensitivity analyses – rationale, strengths and limitations 54 6.6 Data sources 55 Table 5. Metadata about data sources and software 56 6.7 Data management 56 6.8 Quality control 58 6.9 Study size and feasibility 59 7. Limitation of the methods | 6. Research methods | 19 |
| 6.3 Setting 21 6.3.1 Context and rationale for definition of time 0 (and other primary time anchors) for entry to the study population 21 6.3.2 Context and rationale for study inclusion criteria: 22 6.3.3 Context and rationale for study exclusion criteria 22 6.4.4 Variables 22 6.4.1 Context and rationale for exposure(s) of interest 22 6.4.2 Context and rationale for outcome(s) of interest 22 6.4.3 Context and rationale for outcome(s) of interest 22 6.4.4 Context and rationale for follow-up 23 Table 1. Operational Definitions of follow-up 23 6.4.4 Context and rationale for covariates (confounding variables and effect modifiers, e.g. risk factors, comorbidities, comedications) 25 6.5 Data analysis 42 6.5.1 Context and rationale for analysis plan 42 Table 3. Primary, secondary, and subgroup analysis specification 42 Table 4. Sensitivity analyses - rationale, strengths and limitations 54 6.6 Data sources 55 6.6.1 Context and rationale for data sources 55 Table 5. Metadata about data sources and software 56 6.7 Data management 56 6.8 Quality control 58 6.9 Study size and feasibility 59 7. Limitation of the methods | 6.1 Study design | 19 |
| 6.3.1 Context and rationale for definition of time 0 (and other primary time anchors) for entry to the study population 21 6.3.2 Context and rationale for study inclusion criteria: 22 6.3.3 Context and rationale for study exclusion criteria 22 6.3.3 Context and rationale for study exclusion criteria 22 6.4.1 Context and rationale for exposure(s) of interest 22 6.4.1 Context and rationale for outcome(s) of interest 22 6.4.2 Context and rationale for follow-up 23 7 able 1. Operational Definitions of follow-up 23 7 able 1. Operational Definitions of follow-up 23 7 able 2. Operational Definitions of Covariates (confounding variables and effect modifiers, e.g. risk factors, comorbidities, comedications) 25 7 able 2. Operational Definitions of Covariates 25 7 able 3. Primary, secondary, and subgroup analysis specification 42 7 able 4. Sensitivity analyses – rationale, strengths and limitations 54 7 able 4. Sensitivity analyses – rationale, strengths and limitations 55 7 able 5. Metadata about data sources 55 7 able 5. Metadata about data sources 36 8 0.6.1 Context and rationale for data sources 36 8 0.8 Quality control 58 8 0.9 Study size and feasibility 59 8 5 1 Limitation of the methods | 6.2 Study design diagrams for the comparison of tirzepatide vs dulaglutide, semaglutide vs sitagliptin, and tirzepatide vs so | emaglutide. 20 |
| 6.3.2 Context and rationale for study inclusion criteria: 6.3.3 Context and rationale for study exclusion criteria 6.3.4 Variables 6.4 Variables 6.4.1 Context and rationale for exposure(s) of interest 6.4.2 Context and rationale for outcome(s) of interest 6.4.2 Context and rationale for follow-up 6.4.4 Context and rationale for lollow-up 6.4.4 Context and rationale for covariates (confounding variables and effect modifiers, e.g. risk factors, comorbidities, comedications) 7 able 2. Operational Definitions of Covariates 6.5 Data analysis 6.5 Data analysis 6.5.1 Context and rationale for analysis plan 7 able 3. Primary, secondary, and subgroup analysis specification 7 able 4. Sensitivity analyses – rationale, strengths and limitations 6.6 Data sources 6.6.1 Context and rationale for data sources 7 able 5. Metadata about data sources and software 6.7 Data management 6.8 Quality control 6.9 Study size and feasibility 7. Limitation of the methods 59 | 6.3 Setting | 21 |
| 6.3.3 Context and rationale for study exclusion criteria 6.4 Variables 6.4.1 Context and rationale for exposure(s) of interest 6.4.2 Context and rationale for outcome(s) of interest 6.4.2 Context and rationale for follow-up 6.4.3 Context and rationale for follow-up 7 able 1. Operational Definitions of follow-up 7 able 2. Operational Definitions of follow-up 7 able 2. Operational Definitions of Covariates 6.5. Data analysis 6.5. Data analysis 6.5.1 Context and rationale for analysis plan 7 able 3. Primary, secondary, and subgroup analysis specification 7 able 4. Sensitivity analyses – rationale, strengths and limitations 6.6 Data sources 6.6.1 Context and rationale for data sources 7 able 5. Metadata about data sources and software 6.8 Quality control 6.9 Study size and feasibility 7. Limitation of the methods | 6.3.1 Context and rationale for definition of time 0 (and other primary time anchors) for entry to the study population | 21 |
| 6.4 Variables 22 6.4.1 Context and rationale for exposure(s) of interest 22 6.4.2 Context and rationale for outcome(s) of interest 22 6.4.3 Context and rationale for follow-up 23 Table 1. Operational Definitions of follow-up 23 6.4.4 Context and rationale for covariates (confounding variables and effect modifiers, e.g. risk factors, comorbidities, comedications) 25 6.5 Deart analysis 42 6.5 Data analysis 42 6.5.1 Context and rationale for analysis plan 42 Table 3. Primary, secondary, and subgroup analysis specification 42 Table 4. Sensitivity analyses – rationale, strengths and limitations 54 6.6 Data sources 55 6.6.1 Context and rationale for data sources 55 Table 5. Metadata about data sources and software 56 6.7 Data management 56 6.8 Quality control 58 6.9 Study size and feasibility 59 7. Limitation of the methods 59 | 6.3.2 Context and rationale for study inclusion criteria: | 22 |
| 6.4.1 Context and rationale for exposure(s) of interest 6.4.2 Context and rationale for outcome(s) of interest 6.4.3 Context and rationale for follow-up 23 Table 1. Operational Definitions of follow-up 6.4.4 Context and rationale for covariates (confounding variables and effect modifiers, e.g. risk factors, comorbidities, comedications) Table 2. Operational Definitions of Covariates 6.5 Data analysis 6.5.1 Context and rationale for analysis plan 7 table 3. Primary, secondary, and subgroup analysis specification 7 table 4. Sensitivity analyses – rationale, strengths and limitations 7 table 5. Metadata about data sources 6.6.1 Context and rationale for data sources 7 table 5. Metadata about data sources and software 7 table 5. Metadata about data sources and software 7 table 5. Study size and feasibility 7 table 5. Study size and feasibility 7 table 4. Sensitivity and feasibility 7 table 5. Metadata about feasibility 7 table 5. Metadata about data sources and feasibility 7 table 5. Study size and feasibility 7 table 5. Metadata about feasibility 7 table 5. Metadata about feasibility 7 table 5. Metadata about feasibility 7 table 5. Metadata feasibility 8 table 7 tabl | 6.3.3 Context and rationale for study exclusion criteria | 22 |
| 6.4.2 Context and rationale for outcome(s) of interest 6.4.3 Context and rationale for follow-up 23 Table 1. Operational Definitions of follow-up 6.4.4 Context and rationale for covariates (confounding variables and effect modifiers, e.g. risk factors, comorbidities, comedications) Table 2. Operational Definitions of Covariates 6.5 Data analysis 6.5 Data analysis 6.5.1 Context and rationale for analysis plan 42 Table 3. Primary, secondary, and subgroup analysis specification 42 Table 4. Sensitivity analyses – rationale, strengths and limitations 54 6.6 Data sources 6.6.1 Context and rationale for data sources Table 5. Metadata about data sources and software 6.7 Data management 6.8 Quality control 6.9 Study size and feasibility 7. Limitation of the methods 59 | 6.4 Variables | 22 |
| 6.4.3 Context and rationale for follow-up Table 1. Operational Definitions of follow-up 6.4.4 Context and rationale for covariates (confounding variables and effect modifiers, e.g. risk factors, comorbidities, comedications) Table 2. Operational Definitions of Covariates 6.5 Data analysis 6.5 Data analysis 6.5.1 Context and rationale for analysis plan 7 able 3. Primary, secondary, and subgroup analysis specification 7 able 4. Sensitivity analyses – rationale, strengths and limitations 7 able 4. Sensitivity analyses – rationale, strengths and limitations 7 able 5. Metadata about data sources 7 able 5. Metadata about data sources and software 7 able 5. Wetadata about data sources and software 7 able 5. Study size and feasibility 7 thimitation of the methods 7 Limitation of the methods | 6.4.1 Context and rationale for exposure(s) of interest | 22 |
| Table 1. Operational Definitions of follow-up 6.4.4 Context and rationale for covariates (confounding variables and effect modifiers, e.g. risk factors, comorbidities, comedications) Table 2. Operational Definitions of Covariates 6.5 Data analysis 6.5.1 Context and rationale for analysis plan 42 Table 3. Primary, secondary, and subgroup analysis specification 42 Table 4. Sensitivity analyses – rationale, strengths and limitations 54 6.6 Data sources 55 6.6.1 Context and rationale for data sources 55 Table 5. Metadata about data sources and software 6.7 Data management 6.8 Quality control 6.9 Study size and feasibility 7. Limitation of the methods 53 24 42 42 53 42 54 55 55 56 6.9 Study size and feasibility 59 | 6.4.2 Context and rationale for outcome(s) of interest | 22 |
| 6.4.4 Context and rationale for covariates (confounding variables and effect modifiers, e.g. risk factors, comorbidities, comedications) Table 2. Operational Definitions of Covariates 6.5 Data analysis 6.5 Data analysis 6.5.1 Context and rationale for analysis plan 7 Table 3. Primary, secondary, and subgroup analysis specification 7 Table 4. Sensitivity analyses – rationale, strengths and limitations 7 Table 5. Metadata about data sources 7 Table 5. Metadata about data sources and software 8 Table 5. Metadata about data sources and software 9 Table 5. Metadata about data sources and | 6.4.3 Context and rationale for follow-up | 23 |
| Table 2. Operational Definitions of Covariates 6.5 Data analysis 6.5.1 Context and rationale for analysis plan 42 Table 3. Primary, secondary, and subgroup analysis specification Table 4. Sensitivity analyses – rationale, strengths and limitations 54 6.6 Data sources 55 6.6.1 Context and rationale for data sources 55 Table 5. Metadata about data sources and software 6.7 Data management 6.8 Quality control 6.9 Study size and feasibility 7. Limitation of the methods 25 42 42 42 42 43 42 | Table 1. Operational Definitions of follow-up | 23 |
| 6.5 Data analysis 6.5.1 Context and rationale for analysis plan 42 Table 3. Primary, secondary, and subgroup analysis specification 42 Table 4. Sensitivity analyses – rationale, strengths and limitations 54 6.6 Data sources 55 6.6.1 Context and rationale for data sources 55 Table 5. Metadata about data sources and software 56 6.7 Data management 6.8 Quality control 6.9 Study size and feasibility 7. Limitation of the methods 59 | 6.4.4 Context and rationale for covariates (confounding variables and effect modifiers, e.g. risk factors, comorbidities, | comedications) 25 |
| 6.5.1 Context and rationale for analysis plan 42 Table 3. Primary, secondary, and subgroup analysis specification 42 Table 4. Sensitivity analyses – rationale, strengths and limitations 54 6.6 Data sources 6.6.1 Context and rationale for data sources 55 Table 5. Metadata about data sources and software 6.7 Data management 6.8 Quality control 6.9 Study size and feasibility 7. Limitation of the methods 59 | Table 2. Operational Definitions of Covariates | 25 |
| Table 3. Primary, secondary, and subgroup analysis specification Table 4. Sensitivity analyses – rationale, strengths and limitations 54 6.6 Data sources 6.6.1 Context and rationale for data sources Table 5. Metadata about data sources and software 56 6.7 Data management 58 6.9 Study size and feasibility 7. Limitation of the methods 42 4 | 6.5 Data analysis | 42 |
| Table 4. Sensitivity analyses – rationale, strengths and limitations 6.6 Data sources 6.6.1 Context and rationale for data sources Table 5. Metadata about data sources and software 6.7 Data management 6.8 Quality control 6.9 Study size and feasibility 7. Limitation of the methods | 6.5.1 Context and rationale for analysis plan | 42 |
| 6.6 Data sources 55 6.6.1 Context and rationale for data sources 55 Table 5. Metadata about data sources and software 56 6.7 Data management 56 6.8 Quality control 59 7. Limitation of the methods 55 75 | Table 3. Primary, secondary, and subgroup analysis specification | 42 |
| 6.6.1 Context and rationale for data sources Table 5. Metadata about data sources and software 56 6.7 Data management 58 6.8 Quality control 59 7. Limitation of the methods 55 7. Limitation of the methods | Table 4. Sensitivity analyses – rationale, strengths and limitations | 54 |
| Table 5. Metadata about data sources and software 56 6.7 Data management 56 6.8 Quality control 58 6.9 Study size and feasibility 59 7. Limitation of the methods 59 | 6.6 Data sources | 55 |
| 6.7 Data management 56 6.8 Quality control 58 6.9 Study size and feasibility 59 7. Limitation of the methods 59 | 6.6.1 Context and rationale for data sources | 55 |
| 6.8 Quality control 58 6.9 Study size and feasibility 59 7. Limitation of the methods 59 | Table 5. Metadata about data sources and software | 56 |
| 6.9 Study size and feasibility 59 <b>7. Limitation of the methods</b> 59 | 6.7 Data management | 56 |
| 7. Limitation of the methods 59 | 6.8 Quality control | 58 |
| | 6.9 Study size and feasibility | 59 |
| 3. Protection of human subjects 59 | 7. Limitation of the methods | 59 |
| | 8. Protection of human subjects | 59 |

| 9. References 10. Appendices | 59<br>61 |
|---|---|
| 1tirzdula, semasita, tirzsema Target Trial Framework, Operational Definitions, and Data Fitness Assessment | 61 |
| 2tirzdula, semasita, tirzsema Code algorithms | 61 |
| 3tirzdula, semasita, tirzsema Flowchart for cohort assembly | 62 |
| 4tirzdula, semasita, tirzsema 1st feasibility assessment | 62 |
| 5tirzdula, semasita, tirzsema 2nd feasibility assessment | 62 |
| 6tirzdula, semasita, tirzsema Balance Assessment - PS Distribution and C-Statistic | 62 |
| 7tirzdula, semasita, tirzsema Balance Assessment - Table 1 | 62 |

### 2. Abstract

This is a non-randomized, non-interventional study that is part of the *Randomized Controlled Trials Duplicated Using Prospective Longitudinal Insurance Claims: Applying Techniques of Epidemiology* (RCT-DUPLICATE) initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to assess the comparative effectiveness of

- 1. Tirzepatide vs dulaglutide.
- 2. Semaglutide vs sitagliptin,
- 3. Tirzepatide vs semaglutide

on cardiovascular outcomes in individuals typically treated in clinical practice who are at low, moderate, and high cardiovascular risk with type 2 diabetes (T2DM) and overweight but might not meet the eligibility criteria of pivotal RCTs for each drug (SUSTAIN-6 and SURPASS-CVOT trials), used to support regulatory approval in patients at cardiovascular risk.<sup>1,2</sup> Although many features of the target trials cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the target trial. Randomization cannot be achieved in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice.

The three database studies will be new-user active-comparative studies, conducted using 3 national United States claims databases, where we compare the effect of semaglutide vs sitagliptin (used as an active comparator placebo proxy), tirzepatide vs dulaglutide, and tirzepatide vs semaglutide on the composite end point of all-cause mortality, myocardial infarction, or stroke. Clinical guidelines during the study period recommended both tirzepatide and semaglutide for the same indications of glucose lowering and weight reduction.

The study will use three data sources: Optum Clinformatics, Merative MarketScan, and Medicare.

Optum: Study period between January 1, 2018 to February 28, 2025.

MarketScan: Study period between January 1, 2018 to December 31, 2023.

Medicare: Study period between January 1, 2018 to December 31, 2020.

## 3. Amendments and updates

| Version date | Version number | Section of protocol | Amendment or update | Reason |
|---|---|---|---|---|
| 10 August,<br>2025 | 2 | 4,<br>5A and 5B,<br>6.2<br>6.4.2<br>6.5.1 | Add composite outcomes that exclude death as a component or single end point from the comparison of injectable | Benchmarking analyses for the emulation of SUSTAIN-6 comparing injectable semaglutide to sitagliptin (a placebo-proxy) revealed disagreement in the comparison of the secondary outcome of all-cause mortality between the database study and trial, potentially due to residual confounding. The results for the primary and other secondary |

| Coronary<br>disease,<br>Cardiomy<br>Valve dis<br>failure, C | This study focuses on an expanded patient population compared to the SUSTAIN-6 trial. Due to concerns about bias, we will view the results of outcomes that include mortality for comparisons of injectable semaglutide with sitagliptin with scepticism. For the comparison of injectable semaglutide vs sitagliptin in an expanded population, we will add and evaluate different composite cardiovascular outcomes which exclude all-cause mortality, e.g. major adverse |
|---|---|
|---|---|

# 4. Rationale and background

The purpose of this protocol is to specify three target trials assessing the comparative effectiveness of

- 1. the dual glucose-dependent insulinotropic polypeptide (GIP) and glucagon-like peptide-1 receptor agonist (GLP-1-RA) tirzepatide vs the GLP-1-RA dulaglutide.
- 2. the GLP-1-RA semaglutide vs the dipeptidyl peptidase-4 (DPP-4) inhibitor sitagliptin (used as an active comparator placebo proxy),
- 3. the GIP and GLP-1-RA tirzepatide vs the GLP-1-RA semaglutide

on major adverse cardiovascular outcomes (MACE), defined as the composite end point of all-cause mortality, myocardial infarction, or stroke in patients typically treated in clinical practice who are at low, moderate, and high cardiovascular risk with type 2 diabetes and overweight who might not have met strict eligibility criteria of the pivotal RCTs SUSTAIN-6 and SURPASS-CVOT. The results for all-cause mortality or composite outcomes that include death will be viewed with scepticism for the comparison of injectable semaglutide vs sitagliptin because a benchmarking database study designed to emulate the SUSTAIN-6 trial using Optum and MarketScan data yielded divergent results for the mortality outcome.

Injectable semaglutide became available on December 5, 2017 under the brand name Ozempic.<sup>3</sup> On January 16, 2020, the approval was expanded to include cardiovascular risk reduction in adults with type 2 diabetes mellitus and known heart disease. On March 28, 2022, Novo Nordisk received FDA approval for a higher-dose semaglutide (2 mg) to provide improved glycemic control for adults with type 2 diabetes mellitus. Meanwhile, semaglutide received its first FDA approval for the treatment of obesity in adults under the brand name Wegovy on June 4, 2021. On December 23, 2022, the approval was extended to include teenagers aged 12 and older. Later, on March 8, 2024, Wegovy was additionally approved for cardiovascular risk reduction in people with overweight or obesity and established cardiovascular disease. On January 28, 2025, Ozempic became the first and only GLP-1-RA approved to reduce the risk of worsening kidney disease and cardiovascular death in adults with Type 2 diabetes and chronic kidney disease.

Sitagliptin was specifically chosen as an active comparator that could proxy for placebo because a major randomized controlled trial on cardiovascular outcomes demonstrated that it does not affect the cardiovascular outcomes under investigation.<sup>4</sup> This contrasts with other DPP4i such as saxagliptin, which has raised concerns regarding potential increased risks of heart failure, <sup>5-8</sup> and linagliptin, which is commonly prescribed for patients with renal impairment because it does not require dose modifications based on kidney function, potentially leading to increased confounding compared to sitagliptin.<sup>9,10</sup> Sodium-glucose Cotransporter-2 (SGLT2) inhibitors would not be a neutral comparator, as they significantly reduce clinically important kidney events, kidney failure, and cardiovascular events.<sup>11-14</sup> Sulfonylureas (SUs), though inexpensive and widely used, are a poor comparator in cardiovascular outcome studies due to their association with hypoglycemia, weight gain, and channeling bias, as they are often prescribed to elderly, lower socioeconomic status patients with higher baseline cardiovascular risk, making direct comparisons to GLP-1-RAs less reliable.<sup>15</sup>

The GIP/GLP-1-RA tirzepatide became available on May 13, 2022, when it was approved to treat type 2 diabetes mellitus. A year later, on November 8, 2023 tirzepatide was approved for chronic weight management in adults with obesity or overweight who also have at least one weight-related comorbid condition, such as hypertension, dyslipidemia, type 2 diabetes mellitus, obstructive sleep apnea, or cardiovascular disease. Later on, on December 20, 2024, tirzepatide was approved to treat moderate to severe obstructive sleep apnea (OSA) in adults with obesity, to be used in combination with a reduced-calorie diet and increased physical activity.

Dulaglutide was approved on September 18, 2014 to improve glycemic control in adults with T2DM. On February 21, 2020 FDA approved dulaglutide to reduce the risk of major adverse cardiovascular events in adults with T2DM who have established CVD or multiple cardiovascular risk factors. In the same year, on March 9, 2020 an additional dosing regimen was approved. Finally, on November 17, 2022, dulaglutide was approved for use in pediatric patients aged 10 years and older.

# **5.** Research question and objectives

# Table 2. Primary and secondary research questions and objectives

# A. Primary research questions and objectives: Tirzepatide vs dulaglutide

| To evaluate the comparative effect of tirzepatide vs dulaglutide on the composite of all-cause |
|---|
| mortality, myocardial infarction, or stroke in patients typically treated in clinical practice who |
| are at low, moderate, and high cardiovascular risk with type 2 diabetes and overweight. |
| We hypothesize that tirzepatide will be non-inferior to dulaglutide at preventing all-cause |
| mortality, myocardial infarction, or stroke in individuals with low, moderate, or high |
| cardiovascular risk, T2DM, and overweight. In addition, superiority to dulaglutide will be tested |
| if non-inferiority is achieved. |
| Individuals typically treated in clinical practice who are at low, moderate, and high |
| cardiovascular risk with T2DM and overweight. |
| Tirzepatide. |
| Dulaglutide. |
| Composite of all-cause mortality, myocardial infarction, or stroke. |
| 1 day after cohort entry date until the first of outcome, disenrollment, end of study period, |
| discontinuation (45 days grace and risk window), switch between the arms, nursing home |
| admission, or start of any other GLP-1-RA. |
| The outcome will be measured from inpatient hospitalizations and death. |
| Hazard ratio. |

# A. Co-primary research questions and objectives: Injectable semaglutide vs sitagliptin

| Objective: | To evaluate the comparative effect of injectable semaglutide vs sitagliptin on the composite |
|---|---|
| | of all-cause mortality, myocardial infarction, or death in patients typically treated in clinical |
| | practice who are at low, moderate, and high cardiovascular risk with type 2 diabetes and |
| | overweight. |
| Hypothesis: | We hypothesize that injectable semaglutide is superior to sitagliptin at preventing all-cause |
| | mortality, myocardial infarction, or stroke in individuals with low, moderate, or high |
| | cardiovascular risk, T2DM, and overweight. Results from this analysis will be viewed with |
| | scepticism in light of a benchmarking database study designed to emulate the SUSTAIN-6 trial |
| | that yielded divergent results for the mortality outcome. |
| Population (mention key inclusion-exclusion | Individuals typically treated in clinical practice who are at low, moderate, and high |
| criteria): | cardiovascular risk with T2DM and overweight. |
| Exposure: | Injectable semaglutide. |
| Comparator: | Sitagliptin. |
| Outcome: | Composite of all-cause mortality, myocardial infarction, or stroke. |
| Time (when follow-up begins and ends): | 1 day after cohort entry date until the first of outcome, disenrollment, end of study period, |
| | discontinuation (45 days grace and risk window), switch between the arms, nursing home |
| | admission, or start of any other GLP-1-RA (including oral semaglutide). |
| Setting: | The outcome will be measured from inpatient hospitalizations and death. |
| Main measure of effect: | Hazard ratio. |

| Objective: | To evaluate the comparative effect of injectable semaglutide vs sitagliptin on the composite |
|---|---|
| | of myocardial infarction or stroke in patients typically treated in clinical practice who are at low, |
| | moderate, and high cardiovascular risk with type 2 diabetes and overweight. |
| Hypothesis: | We hypothesize that injectable semaglutide is superior to sitagliptin at preventing myocardial |
| | infarction or stroke in individuals with low, moderate, or high cardiovascular risk, T2DM, and |
| | overweight. |
| Population (mention key inclusion-exclusion | Individuals typically treated in clinical practice who are at low, moderate, and high |
| criteria): | cardiovascular risk with T2DM and overweight. |
| Exposure: | Injectable semaglutide. |
| Comparator: | Sitagliptin. |
| Outcome: | Composite of myocardial infarction or stroke. |
| Time (when follow-up begins and ends): | 1 day after cohort entry date until the first of outcome, disenrollment, end of study period, |
| | discontinuation (45 days grace and risk window), switch between the arms, nursing home |
| | admission, or start of any other GLP-1-RA (including oral semaglutide). |
| Setting: | The outcome will be measured from inpatient hospitalizations. |
| Main measure of effect: | Hazard ratio. |

# A. Primary research questions and objectives: Tirzepatide vs injectable semaglutide

| To evaluate the comparative effect of tirzepatide vs semaglutide on the composite of all- |
|---|
| cause mortality, myocardial infarction, or stroke in patients typically treated in clinical practice |
| who are at low, moderate, and high cardiovascular risk with type 2 diabetes and overweight. |
| We hypothesize that tirzepatide will be non-inferior to semaglutide at preventing all-cause |
| mortality, myocardial infarction, or stroke in individuals with low, moderate, or high |
| cardiovascular risk, T2DM, and overweight. In addition, superiority to semaglutide will be |
| tested if non-inferiority is achieved. |
| Individuals typically treated in clinical practice who are at low, moderate, and high |
| cardiovascular risk with T2DM and overweight. |
| Tirzepatide. |
| Injectable semaglutide. |
| Composite of all-cause mortality, myocardial infarction, or stroke. |
| 1 day after cohort entry date until the first of outcome, disenrollment, end of study period, |
| discontinuation (45 days grace and risk window), switch between the arms, nursing home |
| admission, or start of any other GLP-1-RA (including oral semaglutide). |
| The outcome will be measured from inpatient hospitalizations and death. |
| Hazard ratio. |

# **B.** Secondary research questions and objectives: Tirzepatide vs dulaglutide

| Objective: | To evaluate the comparative effect of tirzepatide vs dulaglutide on the individual components of the primary endpoint, i.e., all-cause mortality, myocardial infarction, or stroke in patients typically treated in clinical practice who are at low, moderate, and high cardiovascular risk with type 2 diabetes and overweight. |
|---|---|
| Hypothesis: | We hypothesize that tirzepatide will be non-inferior to dulaglutide at preventing all-cause mortality, myocardial infarction, or stroke in individuals with low, moderate, or high cardiovascular risk, T2DM, and overweight. In addition, superiority to dulaglutide will be tested if non-inferiority is achieved. |
| Population (mention key inclusion-exclusion criteria): | Individuals typically treated in clinical practice who are at low, moderate, and high cardiovascular risk with T2DM and overweight. |
| Exposure: | Tirzepatide. |
| Comparator: | Dulaglutide. |
| Outcome: | Individual components of the primary endpoint, i.e., all-cause mortality, myocardial infarction, or stroke. |

| Time (when follow-up begins and ends): | 1 day after cohort entry date until the first of outcome, disenrollment, end of study period, |
|---|---|
| | discontinuation (45 days grace and risk window), switch between the arms, nursing home |
| | admission, or start of any other GLP-1-RA. |
| Setting: | The outcome will be measured from inpatient hospitalizations and death. |
| Main measure of effect: | Hazard ratio. |

| Objective: | To evaluate the comparative effect of tirzepatide vs dulaglutide on all-cause mortality, |
|---|---|
| | hospitalization for heart failure, or urgent heart failure visits in patients typically treated in |
| | clinical practice who are at low, moderate, and high cardiovascular risk with type 2 diabetes |
| | and overweight. |
| Hypothesis: | We hypothesize that tirzepatide will be non-inferior to dulaglutide at preventing all-cause |
| | mortality and total heart failure events requiring hospitalization and/or urgent heart failure |
| | visits in individuals with low, moderate, or high cardiovascular risk, T2DM, and overweight. In |
| | addition, superiority to dulaglutide will be tested if non-inferiority is achieved. |
| Population (mention key inclusion-exclusion | Individuals typically treated in clinical practice who are at low, moderate, and high |
| criteria): | cardiovascular risk with T2DM and overweight. |
| Exposure: | Tirzepatide. |
| Comparator: | Dulaglutide. |
| Outcome: | Composite of all-cause mortality, hospitalization for heart failure, or urgent heart failure visits |
| | requiring intravenous diuretics. |
| Time (when follow-up begins and ends): | 1 day after cohort entry date until the first of outcome, disenrollment, end of study period, |
| | discontinuation (45 days grace and risk window), switch between the arms, nursing home |
| | admission, or start of any other GLP-1-RA. |
| Setting: | The outcome will be measured from inpatient hospitalizations, intravenous diuretic therapy in |
| | an outpatient setting, and death. |
| Main measure of effect: | Hazard ratio. |

| | To evaluate the comparative effect of tirzepatide vs dulaglutide on the safety outcome of urinary tract infections in patients typically treated in clinical practice who are at low, moderate, and high cardiovascular risk with type 2 diabetes and overweight. |
|---|---|
| Hypothesis: | We hypothesize that tirzepatide will not have a different effect from dulaglutide. |
| Population (mention key inclusion-exclusion | Individuals typically treated in clinical practice who are at low, moderate, and high |
| criteria): | cardiovascular risk with T2DM and overweight. |
| Exposure: | Tirzepatide. |

| Comparator: | Dulaglutide. |
|---|---|
| Outcome: | Urinary tract infections. |
| Time (when follow-up begins and ends): | 1 day after cohort entry date until the first of outcome, disenrollment, end of study period, |
| | discontinuation (45 days grace and risk window), switch between the arms, nursing home |
| | admission, or start of any other GLP-1-RA. |
| Setting: | The outcome will be measured using diagnosis codes in an inpatient or outpatient setting that |
| | are followed by an antibiotic prescription within 7 days of the diagnosis code. |
| Main measure of effect: | Hazard ratio. |

| Objective: | To evaluate the comparative effect of tirzepatide vs dulaglutide on the safety outcome of |
|---|---|
| | serious bacterial infections in patients typically treated in clinical practice who are at low, |
| | moderate, and high cardiovascular risk with type 2 diabetes and overweight. |
| Hypothesis: | We hypothesize that tirzepatide will not have a different effect from dulaglutide. |
| Population (mention key inclusion-exclusion | Individuals typically treated in clinical practice who are at low, moderate, and high |
| criteria): | cardiovascular risk with T2DM and overweight. |
| Exposure: | Tirzepatide. |
| Comparator: | Dulaglutide. |
| Outcome: | Serious bacterial infections. |
| Time (when follow-up begins and ends): | 1 day after cohort entry date until the first of outcome, disenrollment, end of study period, discontinuation (45 days grace and risk window), switch between the arms, nursing home admission, or start of any other GLP-1-RA. |
| Setting: | The outcome will be measured using primary diagnosis codes in an inpatient setting. |
| Main measure of effect: | Hazard ratio. |

| | To evaluate the comparative effect of tirzepatide vs dulaglutide on the safety outcome of gastrointestinal adverse events in patients typically treated in clinical practice who are at low, |
|---|---|
| | moderate, and high cardiovascular risk with type 2 diabetes and overweight. |
| | We hypothesize that tirzepatide will not have more events compared to dulaglutide. |
| Population (mention key inclusion-exclusion | Individuals typically treated in clinical practice who are at low, moderate, and high |
| criteria): | cardiovascular risk with T2DM and overweight. |
| Exposure: | Tirzepatide. |
| Comparator: | Dulaglutide. |
| Outcome: | Gastrointestinal adverse events. |

| Time (when follow-up begins and ends): | 1 day after cohort entry date until the first of outcome, disenrollment, end of study period, |
|---|---|
| | discontinuation (45 days grace and risk window), switch between the arms, nursing home |
| | admission, or start of any other GLP-1-RA. |
| Setting: | The outcome will be measured using diagnosis codes in an inpatient and outpatient setting. |
| Main measure of effect: | Hazard ratio. |

| To evaluate the effect of tirzepatide vs dulaglutide on negative control outcomes, (1) hernia |
|---|
| and (2) lumbar radiculopathy in patients typically treated in clinical practice who are at low, |
| moderate, and high cardiovascular risk with type 2 diabetes and overweight. |
| We hypothesize that tirzepatide will not have a different effect from dulaglutide. |
| Individuals typically treated in clinical practice who are at low, moderate, and high |
| cardiovascular risk with T2DM and overweight. In addition, patients will be excluded with |
| recent hernia or lumbar radiculopathy prior to the follow-up time window (45 days) when |
| studying the negative outcome hernia or lumbar radiculopathy, respectively. |
| Tirzepatide. |
| Dulaglutide. |
| Separate analyses for hernia and lumbar radiculopathy. |
| 1 day after cohort entry date until the first of outcome, disenrollment, end of study period, |
| discontinuation (45 days grace and risk window), switch between the arms, nursing home |
| admission, or start of any other GLP-1-RA. |
| The outcome will be measured using diagnosis codes in an inpatient or outpatient setting. |
| Hazard ratio. |

# **B.** Secondary research questions and objectives: Injectable semaglutide vs sitagliptin

| Objective: | To evaluate the comparative effect of injectable semaglutide vs sitagliptin on the individual components of the primary endpoint, i.e., all-cause mortality, myocardial infarction or stroke in patients typically treated in clinical practice who are at low, moderate, and high cardiovascular risk with type 2 diabetes and overweight. |
|---|---|
| Hypothesis: | We hypothesize that injectable semaglutide will be superior to sitagliptin at preventing myocardial infarction or stroke in individuals with low, moderate, or high cardiovascular risk, T2DM, and overweight. Results from the individual end point of all-cause mortality will be |

| | viewed with scepticism in light of a benchmarking database study designed to emulate the |
|---|---|
| | SUSTAIN-6 trial that yielded divergent results for the mortality outcome. |
| Population (mention key inclusion-exclusion | Individuals typically treated in clinical practice who are at low, moderate, and high |
| criteria): | cardiovascular risk with T2DM and overweight. |
| Exposure: | Injectable semaglutide. |
| Comparator: | Sitagliptin. |
| Outcome: | Individual components of the primary endpoint, i.e., myocardial infarction or stroke. |
| Time (when follow-up begins and ends): | 1 day after cohort entry date until the first of outcome, disenrollment, end of study period, |
| | discontinuation (45 days grace and risk window), switch between the arms, nursing home |
| | admission, or start of any other GLP-1-RA (including oral semaglutide). |
| Setting: | The outcome will be measured from inpatient hospitalizations. |
| Main measure of effect: | Hazard ratio. |

| Objective: | To evaluate the comparative effect of injectable semaglutide vs sitagliptin on all-cause |
|---|---|
| | mortality, hospitalization for heart failure, or urgent heart failure visits in patients typically |
| | treated in clinical practice who are at low, moderate, and high cardiovascular risk with type 2 |
| | diabetes and overweight. |
| Hypothesis: | We hypothesize that injectable semaglutide will be superior to sitagliptin at preventing all- |
| | cause mortality and total heart failure events requiring hospitalization and/or urgent heart |
| | failure visits in individuals with low, moderate, or high cardiovascular risk, T2DM, and |
| | overweight. Results from this analysis will be viewed with scepticism in light of a |
| | benchmarking database study designed to emulate the SUSTAIN-6 trial that yielded divergent |
| | results for the mortality outcome. |
| Population (mention key inclusion-exclusion | Individuals typically treated in clinical practice who are at low, moderate, and high |
| criteria): | cardiovascular risk with T2DM and overweight. |
| Exposure: | Injectable semaglutide. |
| Comparator: | Sitagliptin. |
| Outcome: | Composite of all-cause mortality, hospitalization for heart failure, or urgent heart failure visits |
| | requiring intravenous diuretics. |
| Time (when follow-up begins and ends): | 1 day after cohort entry date until the first of outcome, disenrollment, end of study period, |
| | discontinuation (45 days grace and risk window), switch between the arms, nursing home |
| | admission, or start of any other GLP-1-RA (including oral semaglutide). |
| Setting: | The outcome will be measured from inpatient hospitalizations, intravenous diuretic therapy in |
| | an outpatient setting, and death. |
| Main measure of effect: | Hazard ratio. |

| Objective: | To evaluate the comparative effect of injectable semaglutide vs sitagliptin on hospitalization |
|---|---|
| | for heart failure or urgent heart failure visits in patients typically treated in clinical practice who |
| | are at low, moderate, and high cardiovascular risk with type 2 diabetes and overweight. |
| Hypothesis: | We hypothesize that injectable semaglutide will be superior to sitagliptin at preventing all- |
| | cause mortality and total heart failure events requiring hospitalization and/or urgent heart |
| | failure visits in individuals with low, moderate, or high cardiovascular risk, T2DM, and |
| | overweight. |
| Population (mention key inclusion-exclusion | Individuals typically treated in clinical practice who are at low, moderate, and high |
| criteria): | cardiovascular risk with T2DM and overweight. |
| Exposure: | Injectable semaglutide. |
| Comparator: | Sitagliptin. |
| Outcome: | Composite of hospitalization for heart failure or urgent heart failure visits requiring |
| | intravenous diuretics. |
| Time (when follow-up begins and ends): | 1 day after cohort entry date until the first of outcome, disenrollment, end of study period, |
| | discontinuation (45 days grace and risk window), switch between the arms, nursing home |
| | admission, or start of any other GLP-1-RA (including oral semaglutide). |
| Setting: | The outcome will be measured from inpatient hospitalizations, intravenous diuretic therapy in |
| | an outpatient setting. |
| Main measure of effect: | Hazard ratio. |

| Objective: | To evaluate the comparative effect of injectable semaglutide vs sitagliptin on the safety |
|---|---|
| | outcome of urinary tract infections in patients typically treated in clinical practice who are at |
| | low, moderate, and high cardiovascular risk with type 2 diabetes and overweight. |
| Hypothesis: | We hypothesize that injectable semaglutide will not have a different effect from sitagliptin. |
| Population (mention key inclusion-exclusion | Individuals typically treated in clinical practice who are at low, moderate, and high |
| criteria): | cardiovascular risk with T2DM and overweight. |
| Exposure: | Injectable semaglutide. |
| Comparator: | Sitagliptin. |
| Outcome: | Urinary tract infections. |
| Time (when follow-up begins and ends): | 1 day after cohort entry date until the first of outcome, disenrollment, end of study period, |
| | discontinuation (45 days grace and risk window), switch between the arms, nursing home |
| | admission, or start of any other GLP-1-RA (including oral semaglutide). |
| Setting: | The outcome will be measured using diagnosis codes in an inpatient or outpatient setting that |
| | are followed by an antibiotic prescription within 7 days of the diagnosis code. |
| Main measure of effect: | Hazard ratio. |

| Objective: | To evaluate the comparative effect of injectable semaglutide vs sitagliptin on the safety |
|---|---|
| | outcome of serious bacterial infections in patients typically treated in clinical practice who are |
| | at low, moderate, and high cardiovascular risk with type 2 diabetes and overweight. |
| Hypothesis: | We hypothesize that injectable semaglutide will not have a different effect from sitagliptin. |
| Population (mention key inclusion-exclusion | Individuals typically treated in clinical practice who are at low, moderate, and high |
| criteria): | cardiovascular risk with T2DM and overweight. |
| Exposure: | Injectable semaglutide. |
| Comparator: | Sitagliptin. |
| Outcome: | Serious bacterial infections. |
| Time (when follow-up begins and ends): | 1 day after cohort entry date until the first of outcome, disenrollment, end of study period, |
| | discontinuation (45 days grace and risk window), switch between the arms, nursing home |
| | admission, or start of any other GLP-1-RA (including oral semaglutide). |
| Setting: | The outcome will be measured using primary diagnosis codes in an inpatient setting. |
| Main measure of effect: | Hazard ratio. |

| Objective: | To evaluate the comparative effect of injectable semaglutide vs sitagliptin on the safety |
|---|---|
| | outcome of gastrointestinal adverse events in patients typically treated in clinical practice wh |
| | are at low, moderate, and high cardiovascular risk with type 2 diabetes and overweight. |
| Hypothesis: | We hypothesize that injectable semaglutide will not have more events compared to sitagliptin. |
| Population (mention key inclusion-exclusion | Individuals typically treated in clinical practice who are at low, moderate, and high |
| criteria): | cardiovascular risk with T2DM and overweight. |
| Exposure: | Injectable semaglutide. |
| Comparator: | Sitagliptin. |
| Outcome: | Gastrointestinal adverse events. |
| Time (when follow-up begins and ends): | 1 day after cohort entry date until the first of outcome, disenrollment, end of study period, |
| | discontinuation (45 days grace and risk window), switch between the arms, nursing home |
| | admission, or start of any other GLP-1-RA (including oral semaglutide). |
| Setting: | The outcome will be measured using diagnosis codes in an inpatient and outpatient setting. |
| Main measure of effect: | Hazard ratio. |

| Objective: | To evaluate the effect of injectable semaglutide vs sitagliptin on negative control outcomes, |
|---|---|
| Objective. | |
| | including (1) hernia and (2) lumbar radiculopathy in patients typically treated in clinical practice |
| | who are at low, moderate, and high cardiovascular risk with type 2 diabetes and overweight. |
| Hypothesis: | We hypothesize that semaglutide will not have a different effect from sitagliptin. |
| Population (mention key inclusion-exclusion | Individuals typically treated in clinical practice who are at low, moderate, and high |
| criteria): | cardiovascular risk with T2DM and overweight. In addition, patients will be excluded with |
| | recent hernia or lumbar radiculopathy prior to the follow-up time window (45 days) when |
| | studying the negative outcome hernia or lumbar radiculopathy, respectively. |
| Exposure: | Injectable semaglutide. |
| Comparator: | Sitagliptin. |
| Outcome: | Separate analyses for hernia and lumbar radiculopathy. |
| Time (when follow-up begins and ends): | 1 day after cohort entry date until the first of outcome, disenrollment, end of study period, |
| | discontinuation (45 days grace and risk window), switch between the arms, nursing home |
| | admission, or start of any other GLP-1-RA (including oral semaglutide). |
| Setting: | The outcome will be measured using diagnosis codes in an inpatient or outpatient setting. |
| Main measure of effect: | Hazard ratio. |

# **B.** Secondary research questions and objectives: Tirzepatide vs injectable semaglutide

| Objective: | To evaluate the comparative effect of tirzepatide vs injectable semaglutide on the individual components of the primary endpoint, i.e., all-cause mortality, myocardial infarction, or stroke in |
|---|---|
| | patients typically treated in clinical practice who are at low, moderate, and high cardiovasc |
| | risk with type 2 diabetes and overweight. |
| Hypothesis: | We hypothesize that tirzepatide will be non-inferior to injectable semaglutide at preventing |
| | cause mortality, myocardial infarction, or stroke in individuals with low, moderate, or high |
| | cardiovascular risk, T2DM, and overweight. In addition, superiority to sitagliptin will be tested if |
| | non-inferiority is achieved. |
| Population (mention key inclusion-exclusion | Individuals typically treated in clinical practice who are at low, moderate, and high |
| criteria): | cardiovascular risk with T2DM and overweight. |
| Exposure: | Tirzepatide. |
| Comparator: | Injectable semaglutide. |
| Outcome: | Individual components of the primary endpoint, i.e., all-cause mortality, myocardial infarction, |
| | or stroke. |
| Time (when follow-up begins and ends): | 1 day after cohort entry date until the first of outcome, disenrollment, end of study period, |
| | discontinuation (45 days grace and risk window), switch between the arms, nursing home |
| | admission, or start of any other GLP-1-RA (including oral semaglutide). |
| Setting: | The outcome will be measured from inpatient hospitalizations and death. |

| Main measure of effect: | Hazard ratio. |
|---|---|
| Objective: | To evaluate the comparative effect of tirzepatide vs injectable semaglutide on all-cause |
| | mortality, hospitalization for heart failure, or urgent heart failure visits in patients typically |
| | treated in clinical practice who are at low, moderate, and high cardiovascular risk with type 2 |
| | diabetes and overweight. |
| Hypothesis: | We hypothesize that tirzepatide will be non-inferior to injectable semaglutide at preventing all- |
| | cause mortality and total heart failure events requiring hospitalization and/or urgent heart |
| | failure visits in individuals with low, moderate, or high cardiovascular risk, T2DM, and |
| | overweight. In addition, superiority to semaglutide will be tested if non-inferiority is achieved. |
| Population (mention key inclusion-exclusion | Individuals typically treated in clinical practice who are at low, moderate, and high |
| criteria): | cardiovascular risk with T2DM and overweight. |
| Exposure: | Tirzepatide. |
| Comparator: | Injectable semaglutide. |
| Outcome: | Composite of all-cause mortality, hospitalization for heart failure, or urgent heart failure visits |
| | requiring intravenous diuretics. |
| Time (when follow-up begins and ends): | 1 day after cohort entry date until the first of outcome, disenrollment, end of study period, |
| | discontinuation (45 days grace and risk window), switch between the arms, nursing home |
| | admission, or start of any other GLP-1-RA (including oral semaglutide). |
| Setting: | The outcome will be measured from inpatient hospitalizations, intravenous diuretic therapy in |
| | an outpatient setting, and death. |
| Main measure of effect: | Hazard ratio. |

| Objective: | To evaluate the comparative effect of tirzepatide vs injectable semaglutide on the safety |
|---|---|
| | outcome of urinary tract infections in patients typically treated in clinical practice who are at |
| | low, moderate, and high cardiovascular risk with type 2 diabetes and overweight. |
| Hypothesis: | We hypothesize that tirzepatide will not have a different effect from injectable semaglutide. |
| Population (mention key inclusion-exclusion | Individuals typically treated in clinical practice who are at low, moderate, and high |
| criteria): | cardiovascular risk with T2DM and overweight. |
| Exposure: | Tirzepatide. |
| Comparator: | Injectable semaglutide. |
| Outcome: | Urinary tract infections. |

| Time (when follow-up begins and ends): | 1 day after cohort entry date until the first of outcome, disenrollment, end of study period, |
|---|---|
| | discontinuation (45 days grace and risk window), switch between the arms, nursing home |
| | admission, or start of any other GLP-1-RA (including oral semaglutide). |
| Setting: | The outcome will be measured using diagnosis codes in an inpatient or outpatient setting that |
| | are followed by an antibiotic prescription within 7 days of the diagnosis code. |
| Main measure of effect: | Hazard ratio. |

| Objective: | To evaluate the comparative effect of tirzepatide vs injectable semaglutide on the safety |
|---|---|
| | outcome of serious bacterial infections in patients typically treated in clinical practice who are |
| | at low, moderate, and high cardiovascular risk with type 2 diabetes and overweight. |
| Hypothesis: | We hypothesize that tirzepatide will not have a different effect from injectable semaglutide. |
| Population (mention key inclusion-exclusion | Individuals typically treated in clinical practice who are at low, moderate, and high |
| criteria): | cardiovascular risk with T2DM and overweight. |
| Exposure: | Tirzepatide. |
| Comparator: | Injectable semaglutide. |
| Outcome: | Serious bacterial infections. |
| Time (when follow-up begins and ends): | 1 day after cohort entry date until the first of outcome, disenrollment, end of study period, |
| | discontinuation (45 days grace and risk window), switch between the arms, nursing home |
| | admission, or start of any other GLP-1-RA (including oral semaglutide). |
| Setting: | The outcome will be measured using primary diagnosis codes in an inpatient setting. |
| Main measure of effect: | Hazard ratio. |

| | To evaluate the comparative effect of tirzepatide vs injectable semaglutide on the safety outcome of gastrointestinal adverse events in patients typically treated in clinical practice who are at low, moderate, and high cardiovascular risk with type 2 diabetes and overweight. |
|---|---|
| Hypothesis: | We hypothesize that tirzepatide will not have a different effect from injectable semaglutide. |
| Population (mention key inclusion-exclusion | Individuals typically treated in clinical practice who are at low, moderate, and high |
| criteria): | cardiovascular risk with T2DM and overweight. |
| Exposure: | Tirzepatide. |
| Comparator: | Injectable semaglutide. |
| Outcome: | Gastrointestinal adverse events. |

| Time (when follow-up begins and ends): | 1 day after cohort entry date until the first of outcome, disenrollment, end of study period, |
|---|---|
| | discontinuation (45 days grace and risk window), switch between the arms, nursing home |
| | admission, or start of any other GLP-1-RA (including oral semaglutide). |
| Setting: | The outcome will be measured using diagnosis codes in an inpatient and outpatient setting. |
| Main measure of effect: | Hazard ratio. |

| To evaluate the effect of tirzepatide vs injectable semaglutide on negative control outcomes, |
|---|
| including (1) hernia and (2) lumbar radiculopathy in patients typically treated in clinical practice |
| who are at low, moderate, and high cardiovascular risk with type 2 diabetes and overweight. |
| We hypothesize that tirzepatide will not have a different effect from injectable semaglutide. |
| Individuals typically treated in clinical practice who are at low, moderate, and high |
| cardiovascular risk with T2DM and overweight. In addition, patients will be excluded with |
| recent hernia or lumbar radiculopathy prior to the follow-up time window (45 days) when |
| studying the negative outcome hernia or lumbar radiculopathy, respectively. |
| Tirzepatide. |
| Injectable semaglutide. |
| Separate analyses for hernia and lumbar radiculopathy. |
| 1 day after cohort entry date until the first of outcome, disenrollment, end of study period, |
| discontinuation (45 days grace and risk window), switch between the arms, nursing home |
| admission, or start of any other GLP-1-RA (including oral semaglutide). |
| The outcome will be measured using diagnosis codes in an inpatient or outpatient setting. |
| Hazard ratio. |

## 6. Research methods

## **6.1 Study design**

**Research design (e.g. cohort, case-control, etc.):** New user active-comparator cohort study.

**Rationale for study design choice:** The new user active-comparator design is a powerful design that may be able to address confounding by indication. It accomplishes this, in large part, through judicious selection of an appropriate active-comparator group. While selection of an appropriate comparator in the design phase is crucial, cohort studies often require additional adjustment of measurable confounders. A common method for adjusting for confounding is via a propensity score.

## **6.2 Study design diagrams** for the comparison of tirzepatide vs dulaglutide, semaglutide vs sitagliptin, and tirzepatide vs semaglutide.

Cohort Entry Date (CED, Day 0) sation of exposure Group (Tirzepatide)] OR nsation of Reference Group (Dulaglutide)] Days [0, 0] dCensoring criteria: · Occurrence of outcomes Disenrollment or use of Pramlintide or any GLP-1-RA except tirzepatide or duladutide · End of study period · 365 days after CED · Discontinuation (45 days grace window and risk-window) · Switch to other GLP-1-RA · Nursing home admission EXCL: Concurrent use of both study drugs Days [0] PRIMARY OUTCOME: Composite of all-cause mortality, myocardial infarction, and stroke

Day 0

Figure 1. Study diagram for the comparison tirzepatide vs dulaglutide.

Figure 2. Study diagram for the comparison semaglutide vs sitagliptin.



\*Results including mortality will be viewed with scepticism in light of a benchmarking database study designed to emulate the SUSTAIN-6 trial that yielded divergent results for the mortality outcome. We therefore also assess the composite outcomes that exclude death as a component.

Figure 3. Study diagram for the comparison tirzepatide vs semaglutide.



## 6.3 Setting

## 6.3.1 Context and rationale for definition of time 0 (and other primary time anchors) for entry to the study population

Time 0 in the database studies was defined to emulate randomization to tirzepatide vs dulaglutide/ semaglutide vs sitagliptin/ tirzepatide vs semaglutide in the trial design. See appendix tables 1<sup>tirzdula, semasita, tirzsema</sup> and 2a<sup>tirzdula, semasita, tirzsema</sup> for operational definitions and detailed code algorithms.

### **6.3.2** Context and rationale for study inclusion criteria:

Study inclusion criteria were defined to reflect clinical routine care settings. See appendix tables 1<sup>tirzdula, semasita, tirzsema</sup> and 2<sup>tirzdula, semasita, tirzsema</sup> for operational definitions and detailed code algorithms. A flowchart of the study cohort assembly is provided in appendices 3<sup>tirzdula, semasita, tirzsema</sup>.

### 6.3.3 Context and rationale for study exclusion criteria

Study exclusion criteria were defined to reflect clinical routine care settings. See appendix tables 1<sup>tirzdula, semasita, tirzsema</sup> and 2<sup>tirzdula, semasita, tirzsema</sup> for operational definitions and detailed code algorithms. A flowchart of the study cohort assembly is provided in appendices 3<sup>tirzdula, semasita, tirzsema</sup>.

#### **6.4 Variables**

#### **6.4.1** Context and rationale for exposure(s) of interest

The exposure and comparator were defined to emulate the agents compared for the trial, tirzepatide vs semaglutide (active-comparator). See appendix tables 1<sup>tirzdula, semasita, tirzsema</sup> and 2<sup>tirzdula, semasita, tirzsema</sup> for operational definitions and detailed code algorithms.

## Algorithm to define duration of exposure effect:

Assuming the effect of the drug lasts for 45 days after the last day's supply, we allow a 45 days gap between the dispensation (grace period) and also add 45 days at the end of the last day's supply (exposure risk window).

#### 6.4.2 Context and rationale for outcome(s) of interest

The primary outcome for the database study was defined as MACE (composite of all-cause mortality, myocardial infarction, or stroke). The results for all-cause mortality or composite outcomes that include death will be viewed with scepticism for the comparison of injectable semaglutide vs sitagliptin because a benchmarking database study designed to emulate the SUSTAIN-6 trial using Optum and MarketScan data yielded divergent results for the mortality outcome. See appendix tables 1<sup>tirzdula, semasita, tirzsema</sup> and 2<sup>tirzdula, semasita, tirzsema</sup> for operational definitions and detailed code algorithms. Optum includes death information from the inpatient discharged dead status, social security death master file, and deaths scraped from obituaries or other sources. MarketScan includes information from the inpatient discharged dead status as well as social security death master file. PPV for myocardial infarction using ICD9 codes was 94%. <sup>19-21</sup> PPV for ischemic stroke using ICD9 codes was 95%. Both of the above ICD9 codes were mapped to ICD10, but no validation study was performed. <sup>22</sup>

Secondary outcomes from the trial that will be evaluated include:

1. Individual components of the primary endpoint, i.e., all-cause mortality, myocardial infarction, or stroke.

- 2. Composite of all-cause mortality, hospitalization for heart failure, or urgent heart failure visits requiring intravenous diuretics.
- 3. For semaglutide vs sitagliptin only:
  - a. A composite outcome of myocardial infarction or stroke.
  - b. A composite of hospitalization for heart failure, or urgent heart failure visits requiring intravenous diuretics.

Safety outcomes of interest include:

- 1. Urinary tract infections.
- 2. Serious bacterial infections.
- Gastrointestinal adverse events.

Control outcomes of interest include:

- 1. Hernia (excluding patients with recent outcome prior to the follow-up time window). This is a negative control outcome where no difference in effect is expected for the three comparative studies.
- 2. Lumbar radiculopathy (excluding patients with recent outcome prior to the follow-up time window). This is a negative control outcome where no difference in effect is expected for the three comparative studies.

#### 6.4.3 Context and rationale for follow-up

Both on-treatment (OT) and intention-to-treat (ITT) analyses will be conducted. Adherence in clinical practice databases is expected to be much worse than in the trial, therefore the OT analysis will be the primary analysis. The OT analysis targets the relative hazard of outcomes while on treatment and may more closely emulate the effect observed in highly adherent trial participants. Both OT and ITT analyses will be conducted with up to 1-year follow-up.

## **Table 1. Operational Definitions of follow-up**

| follow-up start | Day 1 | |
|-----------------|-----------------------------|---------|
| follow-up end¹ | Select<br>all that<br>apply | Specify |
| Date of outcome | Yes | |

| Date of death | Yes | Part of the primary outcome. |
|---|---|---|
| End of observation in data | Yes | Date of disenrollment. |
| <b>Day X following index date</b> (specify day) | Yes | Day 365. |
| <b>End of study period</b> (specify date) | Yes | Tirzepatide vs dulaglutide: Different dates for different databases (Optum: February 28, 2025; MarketScan: December 31, 2023). Semaglutide vs sitagliptin: Dates for different databases (Optum: February 2,8 2025, MarketScan December 31, 2023, Medicare December 31, 2020) Tirzepatide vs semaglutide: Different dates for different databases (Optum: February 28, 2025; MarketScan: December 31, 2023). |
| End of exposure (specify operational details, e.g. stockpiling algorithm, grace period) | Yes | 45 days grace window and 45 days risk window. |
| Date of add to/switch from exposure (specify algorithm) | Yes | Date of augmentation or switching from an exposure to a comparator and vice versa. |
| Other date (specify) | Yes | Tirzepatide vs dulaglutide: Censor upon nursing home admission or starting any other GLP-1-RA. Semaglutide vs sitagliptin: Censor upon nursing home admission or starting any other GLP-1-RA (including oral semaglutide) or DPP4i. Tirzepatide vs semaglutide: Censor upon nursing home admission or starting any other GLP-1-RA (including oral semaglutide). |

 $<sup>^{\</sup>rm 1}$  follow-up ends at the first occurrence of any of the selected criteria that end follow-up.

## 6.4.4 Context and rationale for covariates (confounding variables and effect modifiers, e.g. risk factors, comorbidities, comedications)

We identified a series of covariates that were likely confounders due to being strong risk factors for the primary outcome that were associated with choice of treatment. These include demographics, disease severity related variables, comorbid conditions, comedications, frailty, healthcare utilization and markers of health seeking behaviour.

**Table 2. Operational Definitions of Covariates** 

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement<br>characteristics<br>/<br>validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Demographics | | | | | | | | | |
| Age | Cohort entry<br>year – year of<br>birth, (last<br>observed<br>value in the<br>baseline) | Continuous | [0, 0] | n/a | n/a | n/a | tirzdula <sup>4</sup> ,<br>semasita <sup>5</sup> ,<br>tirzsema <sup>6</sup> | n/a | n/a |
| Gender | Male, Female<br>(last observed<br>value in the<br>baseline) | Categorical | [0, 0] | n/a | n/a | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | n/a |
| Race* | White, Black,<br>Other (Asian,<br>Hispanic),<br>Missing/Unkn<br>own (last<br>observed<br>value in the<br>baseline) | Categorical | [0, 0] | n/a | n/a | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | n/a |
| Region | Northeast,<br>Midwest/Nort<br>h central,<br>South, West<br>(last observed<br>value in the<br>baseline) | Categorical | [0, 0] | n/a | n/a | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | n/a |


| Characteristics | Details | Type of<br>variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics / validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Number of antidiabetic drugs on CED | | Continuous | [0, 0] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Concomitant use or initiation of metformin | | Binary | [0, 0] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Concomitant use or initiation of insulin | | Binary | [0, 0] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Concomitant use or initiation of sulfonylureas | | Binary | [0, 0] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Concomitant use or initiation of DPP4i | | Binary | [0, 0] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Concomitant use or initiation of SGLT2i | | Binary | [0, 0] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Concomitant use or initiation of other glucose-lowering drugs | | Binary | [0, 0] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Past use of metformin | | Binary | [-365, -1] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Past use of insulin | | Binary | [-365, -1] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Characteristics | Details | Type of<br>variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement<br>characteristics<br>/<br>validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Past use of sulfonylureas | | Binary | [-365, -1] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Past use of DPP4i | | Binary | [-365, -1] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Past use of SGLT2i | | Binary | [-365, -1] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Past use of other glucose-lowering drugs | | Binary | [-365, -1] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Heart failure medic | ations | | <u> </u> | | | • | | | |
| ACEi / ARB | | Binary | [-365, 0] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| ARNI | | Binary | [-365, 0] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Thiazides | | Binary | [-365, 0] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Beta-blockers | | Binary | [-365, 0] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Calcium channel blockers | | Binary | [-365, 0] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Digoxin / Digitoxin | | Binary | [-365, 0] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics / validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Loop diuretics | | Binary | [-365, 0] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Other diuretics | | Binary | [-365, 0] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Intravenous<br>diuretics | | Binary | [-365, 0] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Nitrates | | Binary | [-365, 0] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Other medications | ; | | | | | | | | |
| Anti-arrhythmics | | Binary | [-365, 0] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Statins | | Binary | [-365, 0] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| PCSK9 inhibitors<br>and other lipid-<br>lowering drugs | | Binary | [-365, 0] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Antiplatelet agents | | Binary | [-365, 0] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Oral<br>anticoagulants | | Binary | [-365, 0] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| COPD/Asthma<br>medication | | Binary | [-365, 0] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of<br>variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics / validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| NSAIDs | | Binary | [-365, 0] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Oral<br>corticosteroids | | Binary | [-365, 0] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Osteoporosis<br>agents (incl.<br>bisphosphonates) | | Binary | [-365, 0] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Opioids | | Binary | [-365, 0] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Anti-depressants | | Binary | [-365, 0] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Antipsychotics | | Binary | [-365, 0] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Anxiolytics/hypnot ics, benzodiazepines | | Binary | [-365, 0] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Medication for dementia | | Binary | [-365, 0] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Urinary tract infections antibiotics | | Binary | [-365, 0] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Laxatives | | Binary | [-365, 0] | n/a | generic | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |

Healthcare utilization markers

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics / validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Number of distinct<br>medications,<br>median (iqr), mean<br>(sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Number of office<br>visits, median (iqr),<br>mean (sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Number of<br>endocrinologist<br>visits, median (iqr),<br>mean (sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Number of<br>cardiologist visits,<br>median (iqr), mean<br>(sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Number of internal<br>medicine/family<br>medicine visits,<br>median (iqr), mean<br>(sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Number of<br>Electrocardiogram<br>s, median (iqr),<br>mean (sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Number of<br>Echocardiograms,<br>median (iqr), mean<br>(sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of<br>variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement<br>characteristics<br>/<br>validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Pharmacy out-of-<br>pocket cost,<br>median (iqr), mean<br>(sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Unique brand<br>medications,<br>median (iqr), mean<br>(sd)** | | Continuous | [-365, 0] | n/a | n/a | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Unique generic<br>medications,<br>median (iqr), mean<br>(sd)** | | Continuous | [-365, 0] | n/a | n/a | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Ratio of unique<br>brand to generic<br>medications,<br>median (iqr), mean<br>(sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Healthy behavior n | narkers | • | | • | | | | | |
| Colonoscopy /<br>Sigmoidoscopy | | Binary | [-365, 0] | Any | CPT/HCPCS | Any | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Flu vaccine /<br>Pneumococcal<br>vaccine | | Binary | [-365, 0] | Any | CPT/HCPCS | Any | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Pap smear test | | Binary | [-365, 0] | Any | CPT/HCPCS | Any | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| PSA test | | Binary | [-365, 0] | Any | CPT/HCPCS | Any | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement<br>characteristics<br>/<br>validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Fecal occult blood test | | Binary | [-365, 0] | Any | CPT/HCPCS | Any | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Bone mineral density tests | | Binary | [-365, 0] | Any | CPT/HCPCS | Any | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Mammograms | | Binary | [-365, 0] | Any | CPT/HCPCS | Any | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Telemedicine | | Binary | [-365, 0] | Any | CPT/HCPCS | Any | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Laboratory and dia | gnostic tests | | | | | | | | |
| Number of HbA1c<br>tests, median (iqr),<br>mean (sd) | | Continuous | [-365, 0] | Any | CPT/HCPCS | Any | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Number of lipid<br>panels, median<br>(iqr), mean (sd) | | Continuous | [-365, 0] | Any | CPT/HCPCS | Any | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Number of<br>creatinine tests,<br>median (iqr), mean<br>(sd) | | Continuous | [-365, 0] | Any | CPT/HCPCS | Any | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Number of<br>natriuretic peptide<br>tests, median (iqr),<br>mean (sd) | | Continuous | [-365, 0] | Any | CPT/HCPCS | Any | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Number of urine<br>tests, median (iqr),<br>mean (sd) | | Continuous | [-365, 0] | Any | CPT/HCPCS | Any | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics / validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Lab values | | | | | | | | | |
| HbA1c** | | Continuous | [-365, 0] | n/a | n/a | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Glucose** | | Continuous | [-365, 0] | n/a | n/a | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Creatinine** | | Continuous | [-365, 0] | n/a | n/a | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Systolic blood pressure** | | Continuous | [-365, 0] | n/a | n/a | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Heart rate** | | Continuous | [-365, 0] | n/a | n/a | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| BMI** | | Continuous | [-365, 0] | n/a | n/a | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| eGFR** | | Continuous | [-365, 0] | n/a | n/a | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| LDL** (mg/dl;<br>mean, sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| HDL** (mg/dl;<br>mean, sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Total cholesterol**<br>(mg/dl; mean, sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of variable | Assessmen t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics / validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Triglyceride**<br>(mg/dl; mean, sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Burden of comorbi | dities | | | | | | | | |
| Combined comorbidity score | | Continuous | [-365, 0] | Any | ICD10-CM | Any | tirzdula,<br>semasita,<br>tirzsema | n/a | Gagne et al.,<br>Sun et al. <sup>23,24</sup> |
| Frailty score | | Continuous | [-365, 0] | Any | ICD10-CM | Any | tirzdula,<br>semasita,<br>tirzsema | n/a | Kim et al. <sup>25</sup> |
| Baseline hospitaliz | ations and hospi | tal metrics | | | | | | | |
| Number of any<br>hospitalization,<br>median (iqr), mean<br>(sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Any hospitalization<br>within prior 91<br>days; n (%) | | Binary | [-91, 0] | n/a | n/a | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Any hospitalization<br>within prior 92-<br>365 days; n (%) | | Binary | [-365, -92] | n/a | n/a | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| 0, 1, >1<br>hospitalizations<br>(any) | | Continuous | [-365, 0] | n/a | n/a | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Hospitalization for heart failure; n (%) | | Binary | [-365, 0] | n/a | n/a | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement<br>characteristics<br>/<br>validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Emergency<br>department visits;<br>n (%) | | Binary | [-365, 0] | n/a | n/a | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Calendar year of co | ohort entry | | | | | | | | |
| 2018 | | Categorical | [0, 0] | n/a | n/a | n/a | semasita | n/a | n/a |
| 2019 | | Categorical | [0, 0] | n/a | n/a | n/a | semasita | n/a | n/a |
| 2020 | | Categorical | [0, 0] | n/a | n/a | n/a | semasita | n/a | n/a |
| 2021 | | Categorical | [0, 0] | n/a | n/a | n/a | semasita | n/a | n/a |
| 2022 | | Categorical | [0, 0] | n/a | n/a | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | n/a |
| 2023 | | Categorical | [0, 0] | n/a | n/a | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | n/a |
| 2024 | | Categorical | [0, 0] | n/a | n/a | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | n/a |
| 2025 | | Categorical | [0, 0] | n/a | n/a | n/a | tirzdula,<br>semasita,<br>tirzsema | n/a | n/a |

<sup>&</sup>lt;sup>1</sup>IP = inpatient, OP = outpatient, ED = emergency department, OT = other, n/a = not applicable

<sup>&</sup>lt;sup>2</sup>See appendix for listing of clinical codes for each study parameter

<sup>&</sup>lt;sup>3</sup> Specify whether a diagnosis code is required to be in the primary position (main reason for encounter)

<sup>&</sup>lt;sup>4</sup>tirzdula = Exposure: Tirzepatide; Reference: Dulaglutide

<sup>&</sup>lt;sup>5</sup>semasita = Exposure: Semaglutide; Reference: Sitagliptin

<sup>&</sup>lt;sup>6</sup>tirzsema = Exposure: Tirzepatide; Reference: Semaglutide

<sup>\*</sup>Available for Optum Clinformatics and Medicare

<sup>\*\*</sup>Not used in the PS model

### 6.5 Data analysis

#### **6.5.1** Context and rationale for analysis plan

The studies will use a propensity score (PS) 1:1 nearest neighbor matching with a caliper of 0.01 on the propensity score scale. The propensity score will be estimated as the probability of initiating tirzepatide vs dulaglutide, semaglutide vs sitagliptin, or tirzepatide vs semaglutide given the baseline patient characteristics using multivariable logistic regression models. As diagnostics for PS models, the study will evaluate distributional covariate balance using standardized differences and c-statistics post-matching. The study will estimate the hazard ratio for injectable tirzepatide vs dulaglutide, semaglutide vs sitagliptin, and tirzepatide vs semaglutide on MACE outcome in the matched population using a Cox proportional hazards model.

Table 3. Primary, secondary, and subgroup analysis specification

#### Primary analysis: Tirzepatide vs dulaglutide

| Hypothesis: | , |
|---|---|
| | patients typically treated in clinical practice who are at low, moderate, and high cardiovascular risk with type 2 |
| | diabetes and overweight. |
| Exposure contrast: | Tirzepatide vs dulaglutide. |
| Outcome: | Composite of all-cause mortality, myocardial infarction, or stroke. |
| Analytic software: | Aetion, SAS 9.4, R.4.4.0, Python 3.13.3 |
| Model(s): | Outcome model: Cox proportional hazards |
| (provide details or code) | Follow-up time * status(0) = exposure |
| Confounding adjustment method | |
| | algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity |
| | score stratification (specify strata definition), other. |
| | 1:1 Propensity score nearest-neighbor matching with a caliper of 0.01 on the propensity score scale. |
| Missing data methods | |
| | imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present. |
| Subgroup Analyses | · |
| | Age <65, Age ≥65, Male, Female, with concomitant SGLT2 inhibitor, without concomitant SGLT2 inhibitor, |
| | individuals at high cardiovascular risk (defined as history of cardiovascular event, coronary/carotid/peripheral |
| | artery revascularization procedure), Coronary heart disease, Cardiomyopathy, Valve disorders, Heart failure, |
| | Concomitant high-intensity lipid-lowering therapy. |

# A. Co-primary analysis: Injectable semaglutide vs sitagliptin

| Hypothesis: | Injectable semaglutide decreases the risk of a composite of all-cause mortality, myocardial infarction, or stroke |
|---|---|
| | in patients typically treated in clinical practice who are at low, moderate, and high cardiovascular risk with type 2 |
| | diabetes and overweight. Results from this analysis will be viewed with scepticism in light of a benchmarking |
| | database study designed to emulate the SUSTAIN-6 trial that yielded divergent results for the mortality |
| | outcome. |
| Exposure contrast: | Injectable semaglutide vs sitagliptin. |
| Outcome: | Composite of all-cause mortality, myocardial infarction, or stroke. |
| Analytic software: | Aetion, SAS 9.4, R.4.4.0, Python 3.13.3 |
| Model(s): | Outcome model: Cox proportional hazards |
| (provide details or code) | Follow-up time * status(0) = exposure |
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score weighting (specify weighting |
| | algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity |
| | score stratification (specify strata definition), other. |
| | 1:1 Propensity score nearest-neighbor matching with a caliper of 0.01 on the propensity score scale. |
| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple |
| | imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present. |
| Subgroup Analyses | List all subgroups |
| | Age <65, Age ≥65, Male, Female, with concomitant SGLT2 inhibitor, without concomitant SGLT2 inhibitor, |
| | individuals at high cardiovascular risk (high cardiovascular risk being defined as having a history of a |
| | cardiovascular event, or coronary, carotid, or peripheral artery revascularization procedure), Coronary heart |
| | disease, Cardiomyopathy, Valve disorders, Heart failure, Concomitant high-intensity lipid-lowering therapy. |
| Hypothesis: | Injectable semaglutide decreases the risk of a composite of myocardial infarction or stroke in patients typically |
| | treated in clinical practice who are at low, moderate, and high cardiovascular risk with type 2 diabetes and |
| F | overweight. |
| Exposure contrast: | Injectable semaglutide vs sitagliptin. |
| Outcome: | Composite of all-cause mortality, myocardial infarction, or stroke. |
| Analytic software: | Aetion, SAS 9.4, R.4.4.0, Python 3.13.3 |
| Model(s): | Outcome model: Cox proportional hazards |
| (provide details or code) | Follow-up time * status(0) = exposure |
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score weighting (specify weighting |
| | algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity |
| | score stratification (specify strata definition), other. |
| _ | 1:1 Propensity score nearest-neighbor matching with a caliper of 0.01 on the propensity score scale. |

| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple |
|---|---|
| | imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present. |
| Subgroup Analyses | List all subgroups |
| | Age <65, Age ≥65, Male, Female, with concomitant SGLT2 inhibitor, without concomitant SGLT2 inhibitor, |
| | individuals at high cardiovascular risk (high cardiovascular risk being defined as having a history of a |
| | cardiovascular event, or coronary, carotid, or peripheral artery revascularization procedure), Coronary heart |
| | disease, Cardiomyopathy, Valve disorders, Heart failure, Concomitant high-intensity lipid-lowering therapy. |

# A. Primary analysis: Tirzepatide vs injectable semaglutide

| Hypothesis: | Tirzepatide does not increase the risk of a composite of death, myocardial infarction, or stroke in patients |
|---|---|
| | typically treated in clinical practice who are at low, moderate, and high cardiovascular risk with type 2 diabetes |
| | and overweight. |
| Exposure contrast: | Tirzepatide vs injectable semaglutide. |
| Outcome: | Composite of all-cause mortality, myocardial infarction, or stroke. |
| Analytic software: | Aetion, SAS 9.4, R.4.4.0, Python 3.13.3 |
| Model(s): | Outcome model: Cox proportional hazards |
| (provide details or code) | Follow-up time * status(0) = exposure |
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score weighting (specify weighting |
| | algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity |
| | score stratification (specify strata definition), other. |
| | 1:1 Propensity score nearest-neighbor matching with a caliper of 0.01 on the propensity score scale. |
| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple |
| | imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present. |
| Subgroup Analyses | List all subgroups |
| | Age <65, Age ≥65, Male, Female, with concomitant SGLT2 inhibitor, without concomitant SGLT2 inhibitor, |
| | individuals at high cardiovascular risk (high cardiovascular risk being defined as having a history of a |
| | cardiovascular event, or coronary, carotid, or peripheral artery revascularization procedure), Coronary heart |
| | disease, Cardiomyopathy, Valve disorders, Heart failure, Concomitant high-intensity lipid-lowering therapy. |

# **Secondary Analyses: Tirzepatide vs dulaglutide**

| Hypothesis: | Tirzepatide vs dulaglutide does not increase the risk of occurrence of the individual components of the primary |
|---|---|
| | endpoint, i.e., all-cause mortality, myocardial infarction, or stroke in patients typically treated in clinical practice |
| | who are at low, moderate, and high cardiovascular risk with type 2 diabetes and overweight. |

| Exposure contrast: | Tirzepatide vs dulaglutide. |
|---|---|
| Outcome: | Individual components of the primary endpoint, i.e., all-cause mortality, myocardial infarction, or stroke. |
| Analytic software: | Aetion, SAS 9.4, R.4.4.0, Python 3.13.3 |
| Model(s): | Outcome model: Cox proportional hazards for all-cause mortality, Aalen-Johansen estimator for myocardial |
| (provide details or code) | infarction and stroke to account for the competing risk of death. |
| | Follow-up time * status(0) = exposure |
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score weighting (specify weighting algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity |
| | score stratification (specify strata definition), other. |
| | 1:1 Propensity score nearest-neighbor matching with a caliper of 0.01 on the propensity score scale. |
| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present. |
| Subgroup Analyses | List all subgroups |
| | N/A. |

| Tirzepatide vs dulaglutide does not increase the risk of occurrence of all-cause deaths and total heart failure |
|---|
| , e e e e e e e e e e e e e e e e e e e |
| events requiring hospitalization and/or urgent heart failure visits in patients typically treated in clinical practice |
| who are at low, moderate, and high cardiovascular risk with type 2 diabetes and overweight. |
| Tirzepatide vs dulaglutide. |
| Composite of all-cause mortality, hospitalization for heart failure, or urgent heart failure visits requiring |
| intravenous diuretics. |
| Aetion, SAS 9.4, R.4.4.0, Python 3.13.3 |
| Outcome model: Cox proportional hazards |
| Follow-up time * status(0) = exposure |
| Name method and provide relevant details, e.g. bivariate, multivariable, propensity score weighting (specify weighting |
| algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity |
| score stratification (specify strata definition), other. |
| 1:1 Propensity score nearest-neighbor matching with a caliper of 0.01 on the propensity score scale. |
| Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple |
| imputation (specify model/variables), other. |
| Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present. |
| List all subgroups |
| N/A. |

| Hypothesis: | Tirzepatide vs dulaglutide has no increased or decreased risk of urinary tract infections (safety outcome) |
|---|---|
| | compared to semaglutide in patients typically treated in clinical practice who are at low, moderate, and high |
| | cardiovascular risk with type 2 diabetes and overweight. |
| Exposure contrast: | Tirzepatide vs dulaglutide. |
| Outcome: | Urinary tract infections. |
| Analytic software: | Aetion, SAS 9.4, R.4.4.0, Python 3.13.3 |
| Model(s): | Outcome model: Cox proportional hazards |
| (provide details or code) | Follow-up time*status(0) = exposure |
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score weighting (specify weighting |
| | algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity |
| | score stratification (specify strata definition), other. |
| | 1:1 Propensity score nearest-neighbor matching with a caliper of 0.01 on the propensity score scale. |
| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple |
| | imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present. |
| Subgroup Analyses | List all subgroups |
| | N/A. |

| Hypothesis: | Tirzepatide vs dulaglutide has no increased or decreased risk of serious bacterial infections (safety outcome) |
|---|---|
| | compared to semaglutide in patients typically treated in clinical practice who are at low, moderate, and high |
| | cardiovascular risk with type 2 diabetes and overweight. |
| Exposure contrast: | Tirzepatide vs dulaglutide. |
| Outcome: | Serious bacterial infections. |
| Analytic software: | Aetion, SAS 9.4, R.4.4.0, Python 3.13.3 |
| Model(s): | Outcome model: Cox proportional hazards |
| (provide details or code) | Follow-up time*status(0) = exposure |
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score weighting (specify weighting |
| | algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity |
| | score stratification (specify strata definition), other. |
| | 1:1 Propensity score nearest-neighbor matching with a caliper of 0.01 on the propensity score scale. |
| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple |
| | imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present. |
| Subgroup Analyses | List all subgroups |
| | N/A. |

| Hypothesis: | Tirzepatide vs dulaglutide has no increased or decreased risk of gastrointestinal adverse events (safety |
|---|---|
| | outcome) compared to semaglutide in patients typically treated in clinical practice who are at low, moderate, |
| | and high cardiovascular risk with type 2 diabetes and overweight. |
| Exposure contrast: | Tirzepatide vs dulaglutide. |
| Outcome: | Gastrointestinal adverse events. |
| Analytic software: | Aetion, SAS 9.4, R.4.4.0, Python 3.13.3 |
| Model(s): | Outcome model: Cox proportional hazards |
| (provide details or code) | Follow-up time*status(0) = exposure |
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score weighting (specify weighting |
| | algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity |
| | score stratification (specify strata definition), other. |
| | 1:1 Propensity score nearest-neighbor matching with a caliper of 0.01 on the propensity score scale. |
| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple |
| | imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present. |
| Subgroup Analyses | List all subgroups |
| | N/A. |

| Hypothesis: | Tirzepatide vs dulaglutide has no effect on risk of negative control outcomes compared to dulaglutide. |
|---|---|
| | Negative control outcomes include (1) hernia and (2) lumbar radiculopathy. |
| Exposure contrast: | Tirzepatide vs dulaglutide. |
| Outcome: | Separate analyses for each negative control outcome, including hernia and lumbar radiculopathy |
| Analytic software: | Aetion, SAS 9.4, R.4.4.0, Python 3.13.3 |
| Model(s): | Outcome model: Cox proportional hazards |
| (provide details or code) | Follow-up time*status(0) = exposure |
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score weighting (specify weighting |
| | algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity score stratification (specify strata definition), other. |
| | 1:1 Propensity score nearest-neighbor matching with a caliper of 0.01 on the propensity score scale. |
| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present. |
| Subgroup Analyses | List all subgroups |
| | N/A. |

# Secondary Analyses: Injectable semaglutide vs sitagliptin

| Hypothesis: | Injectable semaglutide vs sitagliptin decreases the risk of occurrence of the individual components of the |
|---|---|
| | primary endpoint, i.e., myocardial infarction or stroke in patients typically treated in clinical practice who are at |
| | low, moderate, and high cardiovascular risk with type 2 diabetes and overweight. |
| Exposure contrast: | Injectable semaglutide vs sitagliptin. |
| Outcome: | Individual components of the primary endpoint, i.e., myocardial infarction or stroke. |
| Analytic software: | Aetion, SAS 9.4, R.4.4.0, Python 3.13.3 |
| Model(s): | Outcome model: Cox proportional hazards for all-cause mortality, Aalen-Johansen estimator for myocardial |
| (provide details or code) | infarction and stroke to account for the competing risk of death. |
| | Follow-up time * status(0) = exposure |
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score weighting (specify weighting |
| | algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity |
| | score stratification (specify strata definition), other. |
| | 1:1 Propensity score nearest-neighbor matching with a caliper of 0.01 on the propensity score scale. |
| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple |
| | imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present. |
| Subgroup Analyses | List all subgroups |
| | N/A. |

| Hypothesis: | Injectable semaglutide vs sitagliptin decreases the risk of occurrence of all-cause deaths and total heart failure |
|---|---|
| | events requiring hospitalization and/or urgent heart failure visits in patients typically treated in clinical practice |
| | who are at low, moderate, and high cardiovascular risk with type 2 diabetes and overweight. |
| Exposure contrast: | Injectable semaglutide vs sitagliptin. |
| Outcome: | Composite of all-cause mortality, hospitalization for heart failure, or urgent heart failure visits requiring |
| | intravenous diuretics. |
| Analytic software: | Aetion, SAS 9.4, R.4.4.0, Python 3.13.3 |
| Model(s): | Outcome model: Cox proportional hazards |
| (provide details or code) | Follow-up time * status(0) = exposure |
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score weighting (specify weighting |
| | algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity |
| | score stratification (specify strata definition), other. |
| | 1:1 Propensity score nearest-neighbor matching with a caliper of 0.01 on the propensity score scale. |
| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple |
| | imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present. |
| Subgroup Analyses | List all subgroups |

| | N/A. |
|---|---|
| Hypothesis: | Injectable semaglutide vs sitagliptin has no increased or decreased risk of urinary tract infections (safety |
| | outcome) compared to semaglutide in patients typically treated in clinical practice who are at low, moderate, |
| | and high cardiovascular risk with type 2 diabetes and overweight. |
| Exposure contrast: | Injectable semaglutide vs sitagliptin. |
| Outcome: | Urinary tract infections. |
| Analytic software: | Aetion, SAS 9.4, R.4.4.0, Python 3.13.3 |
| Model(s): | Outcome model: Cox proportional hazards |
| (provide details or code) | Follow-up time*status(0) = exposure |
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score weighting (specify weighting |
| | algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity |
| | score stratification (specify strata definition), other. |
| | 1:1 Propensity score nearest-neighbor matching with a caliper of 0.01 on the propensity score scale. |
| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple |
| | imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present. |
| Subgroup Analyses | List all subgroups |
| | N/A. |

| Hypothesis: | , |
|---|---|
| | outcome) compared to semaglutide in patients typically treated in clinical practice who are at low, moderate, |
| | and high cardiovascular risk with type 2 diabetes and overweight. |
| Exposure contrast: | Injectable semaglutide vs sitagliptin. |
| Outcome: | Serious bacterial infections. |
| Analytic software: | Aetion, SAS 9.4, R.4.4.0, Python 3.13.3 |
| Model(s): | Outcome model: Cox proportional hazards |
| (provide details or code) | Follow-up time*status(0) = exposure |
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score weighting (specify weighting |
| | algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity |
| | score stratification (specify strata definition), other. |
| | 1:1 Propensity score nearest-neighbor matching with a caliper of 0.01 on the propensity score scale. |
| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple |
| | imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present. |

| Subgroup Analyses | List all subgroups |
|-------------------|--------------------|
| | N/A. |

| Hypothesis: | Injectable semaglutide vs sitagliptin has no increased or decreased risk of gastrointestinal adverse events |
|---|---|
| | (safety outcome) compared to semaglutide in patients typically treated in clinical practice who are at low, |
| | moderate, and high cardiovascular risk with type 2 diabetes and overweight. |
| Exposure contrast: | Injectable semaglutide vs sitagliptin. |
| Outcome: | Gastrointestinal adverse events. |
| Analytic software: | Aetion, SAS 9.4, R.4.4.0, Python 3.13.3 |
| Model(s): | Outcome model: Cox proportional hazards |
| (provide details or code) | Follow-up time*status(0) = exposure |
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score weighting (specify weighting |
| | algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity |
| | score stratification (specify strata definition), other. |
| | 1:1 Propensity score nearest-neighbor matching with a caliper of 0.01 on the propensity score scale. |
| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple |
| | imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present. |
| Subgroup Analyses | List all subgroups |
| | N/A. |

| Hypothesis: | Injectable semaglutide vs sitagliptin has no effect on risk of negative control outcomes compared to |
|---|---|
| | dulaglutide. Negative control outcomes include (1) hernia and (2) lumbar radiculopathy. |
| Exposure contrast: | Injectable semaglutide vs sitagliptin. |
| Outcome: | Separate analyses for each negative control outcome, including hernia and lumbar radiculopathy |
| Analytic software: | Aetion, SAS 9.4, R.4.4.0, Python 3.13.3 |
| Model(s): | Outcome model: Cox proportional hazards |
| (provide details or code) | Follow-up time*status(0) = exposure |
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score weighting (specify weighting |
| | algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity |
| | score stratification (specify strata definition), other. |
| | 1:1 Propensity score nearest-neighbor matching with a caliper of 0.01 on the propensity score scale. |
| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple |
| | imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present. |

| Subgroup Analyses | List all subgroups |
|-------------------|--------------------|
| | N/A. |

# **Secondary Analyses: Tirzepatide vs injectable semaglutide**

| _ | |
|---|---|
| Hypothesis: | Tirzepatide vs injectable semaglutide does not increase the risk of occurrence of the individual components of |
| | the primary endpoint, i.e., all-cause mortality, myocardial infarction, or stroke in patients typically treated in |
| | clinical practice who are at low, moderate, and high cardiovascular risk with type 2 diabetes and overweight. |
| Exposure contrast: | Tirzepatide vs injectable semaglutide. |
| Outcome: | Individual components of the primary endpoint, i.e., all-cause mortality, myocardial infarction, or stroke. |
| Analytic software: | Aetion, SAS 9.4, R.4.4.0, Python 3.13.3 |
| Model(s): | Outcome model: Cox proportional hazards for all-cause mortality, Aalen-Johansen estimator for myocardial |
| (provide details or code) | infarction and stroke to account for the competing risk of death. |
| | Follow-up time * status(0) = exposure |
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score weighting (specify weighting |
| | algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity |
| | score stratification (specify strata definition), other. |
| | 1:1 Propensity score nearest-neighbor matching with a caliper of 0.01 on the propensity score scale. |
| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple |
| | imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present. |
| Subgroup Analyses | List all subgroups |
| | Age <65, Age ≥65, Male, Female, with concomitant SGLT2 inhibitor, without concomitant SGLT2 inhibitor, |
| | individuals at high cardiovascular risk (defined as history of cardiovascular event, coronary/carotid/peripheral artery revascularization procedure). |
| Hypothesis: | Tirzepatide vs injectable semaglutide does not increase the risk of occurrence of all-cause deaths and total |
| | heart failure events requiring hospitalization and/or urgent heart failure visits in patients typically treated in |
| | clinical practice who are at low, moderate, and high cardiovascular risk with type 2 diabetes and overweight. |
| Exposure contrast: | Tirzepatide vs injectable semaglutide. |
| Outcome: | Composite of all-cause mortality, hospitalization for heart failure, or urgent heart failure visits requiring |
| | intravenous diuretics. |
| Analytic software: | Aetion, SAS 9.4, R.4.4.0, Python 3.13.3 |
| Model(s): | Outcome model: Cox proportional hazards |
| (provide details or code) | Follow-up time * status(0) = exposure |

| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score weighting (specify weighting |
|---|---|
| | algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity |
| | score stratification (specify strata definition), other. |
| | 1:1 Propensity score nearest-neighbor matching with a caliper of 0.01 on the propensity score scale. |
| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple |
| | imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present. |
| Subgroup Analyses | List all subgroups |
| | N/A. |

| Hypothesis: | Tirzepatide vs injectable semaglutide has no increased or decreased risk of urinary tract infections (safety |
|---|---|
| | outcome) compared to semaglutide in patients typically treated in clinical practice who are at low, moderate, |
| | and high cardiovascular risk with type 2 diabetes and overweight. |
| Exposure contrast: | Tirzepatide vs injectable semaglutide. |
| Outcome: | Urinary tract infections. |
| Analytic software: | Aetion, SAS 9.4, R.4.4.0, Python 3.13.3 |
| Model(s): | Outcome model: Cox proportional hazards |
| (provide details or code) | Follow-up time*status(0) = exposure |
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score weighting (specify weighting |
| | algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity |
| | score stratification (specify strata definition), other. |
| | 1:1 Propensity score nearest-neighbor matching with a caliper of 0.01 on the propensity score scale. |
| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple |
| | imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present. |
| Subgroup Analyses | List all subgroups |
| | N/A. |

| Hypothesis: | Tirzepatide vs injectable semaglutide has no increased or decreased risk of serious bacterial infections (safety outcome) compared to semaglutide in patients typically treated in clinical practice who are at low, moderate, and high cardiovascular risk with type 2 diabetes and overweight. |
|---|---|
| Exposure contrast: | Tirzepatide vs injectable semaglutide. |
| Outcome: | Serious bacterial infections. |
| Analytic software: | Aetion, SAS 9.4, R.4.4.0, Python 3.13.3 |
| Model(s): | Outcome model: Cox proportional hazards |

| (provide details or code) | Follow-up time*status(0) = exposure |
|---|---|
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score weighting (specify weighting |
| | algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity |
| | score stratification (specify strata definition), other. |
| | 1:1 Propensity score nearest-neighbor matching with a caliper of 0.01 on the propensity score scale. |
| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple |
| | imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present. |
| Subgroup Analyses | List all subgroups |
| | N/A. |

| Hypothesis: | Tirzepatide vs injectable semaglutide has no increased or decreased risk of gastrointestinal adverse events |
|---|---|
| | (safety outcome) compared to semaglutide in patients typically treated in clinical practice who are at low, |
| | moderate, and high cardiovascular risk with type 2 diabetes and overweight. |
| Exposure contrast: | Tirzepatide vs injectable semaglutide. |
| Outcome: | Gastrointestinal adverse events. |
| Analytic software: | Aetion, SAS 9.4, R.4.4.0, Python 3.13.3 |
| Model(s): | Outcome model: Cox proportional hazards |
| (provide details or code) | Follow-up time*status(0) = exposure |
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score weighting (specify weighting |
| | algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity |
| | score stratification (specify strata definition), other. |
| | 1:1 Propensity score nearest-neighbor matching with a caliper of 0.01 on the propensity score scale. |
| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple |
| | imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present. |
| Subgroup Analyses | List all subgroups |
| | N/A. |

| Hypothesis: | Tirzepatide vs injectable semaglutide has no effect on risk of negative control outcomes compared to |
|---|---|
| | dulaglutide. Negative control outcomes include (1) hernia and (2) lumbar radiculopathy. |
| Exposure contrast: | Tirzepatide vs injectable semaglutide. |
| Outcome: | Separate analyses for each negative control outcome, including hernia and lumbar radiculopathy |
| Analytic software: | Aetion, SAS 9.4, R.4.4.0, Python 3.13.3 |
| Model(s): | Outcome model: Cox proportional hazards |

| (provide details or code) | Follow-up time*status(0) = exposure |
|---|---|
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score weighting (specify weighting |
| | algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity |
| | score stratification (specify strata definition), other. |
| | 1:1 Propensity score nearest-neighbor matching with a caliper of 0.01 on the propensity score scale. |
| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple |
| | imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present. |
| Subgroup Analyses | List all subgroups |
| | N/A. |

 Table 4. Sensitivity analyses – rationale, strengths and limitations

| | What is being varied? How? | Why?<br>(What do you expect to<br>learn?) | Strengths of the sensitivity analysis compared to the primary | Limitations of the sensitivity analysis compared to the primary |
|---|---|---|---|---|
| Negative control outcomes, including hernia and lumbar radiculopathy | We evaluate negative control outcomes of hernia and lumbar radiculopathy, where no causal effect is expected from tirzepatide, dulaglutide, semaglutide, or sitagliptin. | We will evaluate the potential impact of residual confounding on this outcome for which there is not expected to be a causal effect | The evaluates the robustness<br>of the interpretation of the<br>primary analysis by evaluating<br>the potential magnitude of<br>unmeasured confounding | This analysis assumes that the confounding structure is the same or similar for the negative control outcome as the outcome of interest |
| Effect estimation in individuals with HbA1c measurement. | The population will be restricted to individuals with a HbA1c measurement in the 120 days before cohort entry. | To assess the impact of restricting to individuals with HbA1c measurement and including HbA1c in the PS model. | Includes baseline glycemic information as captured in laboratory HbA1c measurements. | This approach highly restricts the number of eligible individuals under study and thereby the statistical power of the analysis. |
| As-started analyses (observational analogue to intention-to-treat) to address potential informative censoring. | To address potential informative censoring. | We will consider the first-<br>used medication for 365<br>days without considering<br>drug discontinuation or<br>switching, mimicking an<br>"intention-to-treat"<br>approach. | Reflects follow-up regimen of RCT. | Persistence of drug use is shorter in clinical practice whereas adherence is typically higher in RCTs. Therefore, we expect the estimated effects will be diluted toward the null, underestimating the true treatment effect had patients remained on therapy. |

#### 6.6 Data sources

#### 6.6.1 Context and rationale for data sources

**Reason for selection:** The studies will be conducted in 3 US health care claims databases: Optum Clinformatics (2018-2025), Merative MarketScan (2018-2023), and Medicare (2018-2020). Data from the Merative MarketScan database will only be included if sufficient sample size can be accrued.

**Strengths of data source(s):** Each data source contains deidentified, longitudinal, date-stamped information on patient enrollment, demographics, inpatient/outpatient diagnosis and procedures, admission and discharge dates, and medication dispensation. The death data is captured in the Optum database from inpatient discharge status, social security death master file, and deaths scraped from obituaries or other sources. The death data in MarketScan is captured from the social security death master file and inpatient discharge status. It is recognized that the social security death master file has high specificity and positive predictive value for deaths. While this data resource has under captured deaths since 2011, the capture of deaths is not expected to be differential between compared exposure groups. The death data is captured in the Medicare database from inpatient discharge status, and social security death master file. <sup>26-28</sup>

Limitations of data source(s): Patient healthcare encounters are only observable when they are enrolled in an insurance plan that contributes to the database. Patients may change insurance plans for multiple reasons. Both Optum Clinformatics and Merative MarketScan are primarily employer based insurance databases where patients may disenroll with job changes. In claims data, dispensing data for inpatient medication is unavailable. Diagnoses reflect billing practices, therefore algorithms (preferably validated) are needed for accurate phenotyping of patient conditions. Services that are not covered by insurance do not appear in the data. The trial evaluated cardiovascular deaths, however we will evaluate all-cause mortality in the emulation because most deaths in this cohort of patients at high cardiovascular risk will be related to cardiovascular reasons, the cause of death is not recorded for databases not linked to NDI, and the performance of NDI at identifying cardiovascular causes of death may be suboptimal. <sup>28</sup>

#### **Data source provenance/curation:**

Information about Optum Clinformatics and Merative MarketScan can be found in data dictionaries and user guides that are provided to clients.

Table 5. Metadata about data sources and software

| | Data 1 | Data 2 | Data 3 |
|---|---|---|---|
| Data Source(s): | Optum Clinformatics | Merative MarketScan | Medicare |
| Study Period: | 13 <sup>th</sup> May 2022 | 13 <sup>th</sup> May 2022 | January 1, 2018 |

| Eligible Cohort Entry Period: | Tirzepatide vs dulaglutide:<br>February 28, 2025 | Tirzepatide vs dulaglutide:<br>December 31, 2023 | Semaglutide vs sitagliptin:<br>December 31, 2020 |
|---|---|---|---|
| | Semaglutide vs sitagliptin:<br>February 28, 2025 | Semaglutide vs sitagliptin:<br>December 31, 2023 | |
| | Tirzepatide vs semaglutide:<br>February 28, 2025 | Tirzepatide vs semaglutide:<br>December 31, 2023 | |
| Data Version (or date of last update): | April 2025 | Mortality Cut Set A<br>Received 2024-03-01 | DUA 59286_Received 2023-10-17 |
| Data sampling/extraction criteria: | n/a | n/a | Patients with a diabetes or heart failure diagnosis |
| Type(s) of data: | Administrative claims | Administrative claims | Administrative healthcare claims |
| Data linkage: | n/a | n/a | Linkage to National Death<br>Index |
| Conversion to CDM*: | n/a | n/a | n/a |
| Software for data management: | Aetion Evidence Platform® (2025) | Aetion Evidence Platform® (2025) | Aetion Evidence Platform® (2025) |

<sup>\*</sup>CDM = Common Data Model

#### **6.7 Data management**

<u>Tracking data:</u> The Data Use Agreement (DUA) Custodian (Principal Investigator) and the Division Operations Manager (Winta Tekle) are responsible for receiving and creating a record of new data associated with the given request. The Operations Manager is responsible for all indexing and archiving of documents and electronic media related to data that the Division receives and will log data location, data contents, and associated DUA and Institutional Review Board (IRB) numbers in the Division's centralized tracking system.

<u>Handling and storage:</u> In-scope data will be stored utilizing Mass General Brigham approved information systems – i.e., Division servers and Mass General Brigham network storage.

<u>Archiving</u>: Data retention and any removal will be executed by the Division Operations Manager (Winta Tekle) and Data Manager (Todd MacGarvey). The Division follows Mass General Brigham enterprise record retention policies and follow the terms of the agreement through which the in-scope data was received.

<u>Information security</u>: The Division follows Mass General Brigham's Enterprise Information Security Program (EISP). The EISP helps by providing assurance that Mass General Brigham information and information systems are protected from unauthorized access, use, disclosure, duplication,

modification, or destruction in order to maintain their confidentiality, integrity, and availability. To that end, the EISP policies, standards and procedures create an information security framework that is aligned with the recommendations of the International Organization for Standardization's (ISO) publication 27001 and the National Institute of Standards and Technology's (NIST) publication 800-53 Family of Controls and MGB regulatory and legal requirements (as a HIPAA covered entity).

Mass General Brigham workforce members are required to complete new workforce privacy and information security training upon hire and annually thereafter. Refresh training is provided as appropriate. Mass General Brigham workforce members are required to review and sign a Confidentiality Agreement upon hire and annually thereafter. Additionally, we follow Enterprise Information Security and Privacy policies, including Managing Workforce Members Information Security Responsibilities Policy, which was developed to help assure that Mass General Brigham workforce members are competent and eligible to support the information security responsibilities associated with their role. Mass General Brigham workforce, including Division staff, are required to comply with Enterprise Information Security and Privacy Policies.

<u>Facilities:</u> The research team uses a highly secure, state-of-the-art, computing facility housed at Mass General Brigham's Corporate Data Centers in Needham and Marlborough, Massachusetts as well as Amazon Web Services (AWS). We maintain redundant storage for maximal data integrity and high-speed data access.

The Division uses Mass General Brigham corporate provisioned servers to analyze and store data in connection with this project. There are strict access controls enforced by technical means to ensure that only study staff who have been approved to conduct data analyses and contracted data engineers are able to access data (e.g., Mass General Brigham Authentication (Active Directory) utilized; auditing, logging, and monitoring enabled; firewalls enabled; etc.). All Division servers used in this study are accessible to only authorized staff only through the MGB network and utilizing VPN as appropriate (i.e., users must be on the network and logged into VPN to access). Mass General Brigham has a network information security monitoring team and in-scope servers are enrolled in enterprise security tools (e.g., vulnerability scanning service, antivirus, etc.).

The Division also uses AWS. In-scope AWS services / resources have undergone review and assessment by Mass General Brigham's Information Security Risk Assessment Team/ InfoSec Risk Management Team as required and in alignment with NIST 800-30: Guide for Conducting Risk Assessments. In-scope AWS servers are for our exclusive use (reserved instances), are covered under our organization's Business Associate Agreement with AWS. In-scope servers are housed in anonymous facilities that are not branded as AWS facilities. Physical access is strictly controlled both at the perimeter and at building ingress points by professional security staff utilizing video surveillance, intrusion detection systems, and other electronic means.

Security attributes and controls for the Division's use of in-scope AWS in connection with this project include: encryption at rest and in transit (industry standard AES-256 encryption, SSL/TSL), anti-malware, latest OS updates and patches as well as anti-virus; multi-factor authentication (MFA), Identity and Access Management, including SSO; auditing and logging; principle of least privilege, including for traffic and ports (e.g., deny all default configurations), use of VPC enabled Step functions, etc.; separation between environments; minimum necessary (out of the box AWS roles are not used as they can be overly permissive); all data would reside in the US domestic regions – use only US east HIPAA compliant region; performance monitoring enabled and reviewed as per internal processes; passwords compliant with enterprise password policy and, as appropriate, more protective password requirements; etc. Our Division's AWS use is also subject to ongoing evaluation and monitoring as well – e.g., vulnerability scanning and management, access review, etc.

A data file list will be maintained in Amazon S3 and tracked through Cloudtrail and Cloudwatch. Reporting of data file availability for any file stored in an S3 bucket will be controlled by MGB.

Amazon EC2, Amazon EBS, and Amazon VPC are integrated with AWS CloudTrail, a service that provides a record of actions taken by a user, role, or an AWS service in Amazon EC2, Amazon EBS, and Amazon VPC. CloudTrail captures all API calls for Amazon EC2, Amazon EBS, and Amazon VPC as events, including calls from the console and from code calls to the APIs. MGB IT/security staff have full access to CloudTrail to ensure that CloudTrail monitoring is available at all times. Amazon CloudWatch Events delivers a near-real-time stream of system events that describe changes in AWS resources. Amazon CloudTrail can log, continuously monitor, and retain account activity related to actions across the MGB AWS infrastructure. CloudTrail provides event history of MGB AWS account activity. This event history simplifies security analysis, resource change tracking, and troubleshooting and complies with requirements to ensure the data file inventory is controlled by MGB.

<u>Backups:</u> Backups are created using industry recognized Cryptographic mechanisms (e.g., 256-bit AES encryption) as appropriate and required. Data are backed up within the MGB network from the MGB Needham data center to the MGB Marlborough data center via replication/mirroring and volume-level snapshots. AWS Backup supports both instance-level backups as Amazon Machine Images (AMIs) and volume-level backups as separate snapshots based on the resource tags. AMIs allow MGB IT and security staff to create backups of all S3 and EC2 instances.

In addition to the safeguards listed above, the Division follows enterprise privacy and information security policies and maintains internally procedures in connection with this project to safeguard the data in connection with this project as appropriate and required including: Physical Security and Environmental Controls for Electronic Information Policy; IT Access Control Standards for Users policy; Safeguarding Fax Copiers Printers Telephone Use and Pagers; Physical Removal and Transport of Protected Health Information and Personal Information policy, etc.

#### **6.8 Quality control**

Senior Programmers and Research Specialists perform QA/QC on raw or common data model converted data via SAS/R/Aetion software. The protocol will be iteratively developed and pre-specified data checks including feasibility counts and balance on baseline covariates will be conducted with outputs reviewed by MGB team members. Team members will review code lists to ensure fidelity to intended algorithms.

#### 6.9 Study size and feasibility

See appendices 4<sup>tirzdula, semasita, tirzsema</sup> and appendices 5<sup>tirzdula, semasita, tirzsema</sup> (feasibility, weighting on age, sex, comorbidity score as well as all predefined propensity score variables). Propensity score distribution plots with c-statistics are available in appendices 6<sup>tirzdula, semasita, tirzsema</sup>. Tables 1<sup>tirzdula, semasita, tirzsema</sup> showing prevalence of baseline characteristics and standardized differences in distribution are available in appendices 7<sup>tirzdula, semasita, tirzsema</sup>. Additional diagnostic evaluations, including balance assessments of laboratory and clinical examination test results not included in the propensity score will be conducted to assess potential residual confounding and divergence of treatment over time.

#### 7. Limitation of the methods

As we are using secondary data and the data were not collected for research purposes, some important variables may not be collected or will be measured imperfectly. We have selected validated algorithms when possible and we have created proxies for important variables that are not directly captured in the data to reduce confounding by unmeasured factors.

Although we plan to emulate the important features of each trial as closely as possible in healthcare claims, there may be some elements of the RCT design that are not emulable with a database study, which means that the real-world evidence obtained from the database study and trial will address slightly different clinical questions. For example, in routine clinical care, adherence to treatment is typically not as high as it is in an RCT with strong measures in place to encourage adherence to the study protocol. This means that there is more discontinuation and short-term medication use in the patients identified in claims databases than trial participants.

Apparent agreement between RCT and database study results could occur if the effects of multiple factors (chance, emulation differences, bias) cancel each other out.

## 8. Protection of human subjects

This study has been approved by the Brigham and Women's Hospital Institutional Review Board.

#### 9. References

- 1. Packer M, Zile MR, Kramer CM, et al. Tirzepatide for Heart Failure with Preserved Ejection Fraction and Obesity. N Engl J Med. 2025;392(5):427-437. doi:10.1056/NEJMoa2410027
- 2. Kosiborod MN, Petrie MC, Borlaug BA, et al. Semaglutide in Patients with Obesity-Related Heart Failure and Type 2 Diabetes. *N Engl J Med*. 2024;390(15):1394-1407. doi:10.1056/NEJMoa2313917
- 3. News Details. Novo Nordisk. Accessed February 17, 2025. https://www.novonordisk.com/content/nncorp/global/en/news-and-media/news-and-ir-materials/news-details.html
- 4. Green JB, Bethel MA, Armstrong PW, et al. Effect of Sitagliptin on Cardiovascular Outcomes in Type 2 Diabetes. *N Engl J Med*. 2015;373(3):232-242. doi:10.1056/NEJMoa1501352
- 5. Scirica BM, Bhatt DL, Braunwald E, et al. Saxagliptin and Cardiovascular Outcomes in Patients with Type 2 Diabetes Mellitus. *N Engl J Med*. 2013;369(14):1317-1326. doi:10.1056/NEJMoa1307684
- 6. Heart Failure, Saxagliptin, and Diabetes Mellitus: Observations from the SAVOR-TIMI 53 Randomized Trial. doi:10.1161/CIRCULATIONAHA.114.010389
- 7. A Multicenter Observational Study of Incretin-based Drugs and Heart Failure | New England Journal of Medicine. Accessed December 2, 2024. https://www-nejmorg.emedien.ub.uni-muenchen.de/doi/10.1056/NEJMoa1506115

- 8. Risk for Hospitalized Heart Failure Among New Users of Saxagliptin, Sitagliptin, and Other Antihyperglycemic Drugs: A Retrospective Cohort Study: Annals of Internal Medicine: Vol 164, No 11. Accessed December 2, 2024. https://www.acpjournals.org/doi/10.7326/M15-2568
- 9. Patorno E, Gopalakrishnan C, Bartels DB, Brodovicz KG, Liu J, Schneeweiss S. Preferential prescribing and utilization trends of diabetes medications among patients with renal impairment: Emerging role of linagliptin and other dipeptidyl peptidase 4 inhibitors. *Endocrinol Diabetes Metab*. 2018;1(1):e00005. doi:10.1002/edm2.5
- 10. Gallwitz B. Safety and efficacy of linagliptin in type 2 diabetes patients with common renal and cardiovascular risk factors. *Ther Adv Endocrinol Metab*. 2013;4(3):95-105. doi:10.1177/2042018813486165
- 11. Anker SD, Butler J, Filippatos G, et al. Empagliflozin in Heart Failure with a Preserved Ejection Fraction. *N Engl J Med*. 2021;385(16):1451-1461. doi:10.1056/NEJMoa2107038
- 12. Packer M, Anker SD, Butler J, et al. Cardiovascular and Renal Outcomes with Empagliflozin in Heart Failure. *N Engl J Med*. 2020;383(15):1413-1424. doi:10.1056/NEJMoa2022190
- 13. McMurray JJV, Solomon SD, Inzucchi SE, et al. Dapagliflozin in Patients with Heart Failure and Reduced Ejection Fraction. N Engl J Med. 2019;381(21):1995-2008. doi:10.1056/NEJMoa1911303
- 14. Solomon SD, McMurray JJV, Claggett B, et al. Dapagliflozin in Heart Failure with Mildly Reduced or Preserved Ejection Fraction. N Engl J Med. 2022;387(12):1089-1098. doi:10.1056/NEJMoa2206286
- 15. Mohan V, Saboo B, Khader J, et al. Position of Sulfonylureas in the Current ERA: Review of National and International Guidelines. *Clin Med Insights Endocrinol Diabetes*. 2022;15:11795514221074663. doi:10.1177/11795514221074663
- 16. FDA approves Lilly's Mounjaro<sup>™</sup> (tirzepatide) injection, the first and only GIP and GLP-1 receptor agonist for the treatment of adults with type 2 diabetes | Eli Lilly and Company. Accessed February 17, 2025. https://investor.lilly.com/news-releases/news-release-details/fda-approves-lillys-mounjarotm-tirzepatide-injection-first-and
- 17. Schneeweiss S. A basic study design for expedited safety signal evaluation based on electronic healthcare data. *Pharmacoepidemiol Drug Saf.* 2010;19(8):858-868. doi:10.1002/pds.1926
- 18. Ray WA. Evaluating medication effects outside of clinical trials: new-user designs. Am J Epidemiol. 2003;158(9):915-920. doi:10.1093/aje/kwg231
- 19. Kiyota Y, Schneeweiss S, Glynn RJ, Cannuscio CC, Avorn J, Solomon DH. Accuracy of medicare claims-based diagnosis of acute myocardial infarction: estimating positive predictive value on the basis of review of hospital records. *Am Heart J*. 2004;148(1):99-104. doi:10.1016/j.ahj.2004.02.013
- 20. Andrade SE, Harrold LR, Tjia J, et al. A systematic review of validated methods for identifying cerebrovascular accident or transient ischemic attack using administrative data. *Pharmacoepidemiol Drug Saf.* 2012;21 Suppl 1(Suppl 1):100-128. doi:10.1002/pds.2312
- 21. Roumie CL, Mitchel E, Gideon PS, Varas-Lorenzo C, Castellsague J, Griffin MR. Validation of ICD-9 codes with a high positive predictive value for incident strokes resulting in hospitalization using Medicaid health data. *Pharmacoepidemiol Drug Saf*. 2008;17(1):20-26. doi:10.1002/pds.1518
- 22. Wahl PM, Rodgers K, Schneeweiss S, et al. Validation of claims-based diagnostic and procedure codes for cardiovascular and gastrointestinal serious adverse events in a commercially-insured population. *Pharmacoepidemiol Drug Saf*. 2010;19(6):596-603. doi:10.1002/pds.1924

- 23. Gagne JJ, Glynn RJ, Avorn J, Levin R, Schneeweiss S. A combined comorbidity score predicted mortality in elderly patients better than existing scores. *J Clin Epidemiol*. 2011;64(7):749-759. doi:10.1016/j.jclinepi.2010.10.004
- 24. Sun JW, Rogers JR, Her Q, et al. Adaptation and Validation of the Combined Comorbidity Score for ICD-10-CM. *Med Care*. 2017;55(12):1046-1051. doi:10.1097/MLR.0000000000000824
- 25. Kim DH, Schneeweiss S, Glynn RJ, Lipsitz LA, Rockwood K, Avorn J. Measuring Frailty in Medicare Data: Development and Validation of a Claims-Based Frailty Index. *J Gerontol A Biol Sci Med Sci*. 2018;73(7):980-987. doi:10.1093/gerona/glx229
- 26. Hill ME, Rosenwaike I. The Social Security Administration's Death Master File: the completeness of death reporting at older ages. Soc Secur Bull. 2001;64(1):45-51.
- 27. Death Information in the Research Identifiable Medicare Data | ResDAC. Accessed December 2, 2024. https://resdac.org/articles/death-information-research-identifiable-medicare-data
- 28. Olubowale OT, Safford MM, Brown TM, et al. Comparison of Expert Adjudicated Coronary Heart Disease and Cardiovascular Disease Mortality With the National Death Index: Results From the REasons for Geographic And Racial Differences in Stroke (REGARDS) Study. *J Am Heart Assoc*. 2017;6(5):e004966. doi:10.1161/JAHA.116.004966

## 10. Appendices

See accompanying excel files that specify the cohort studies (tirzdula = Exposure: Tirzepatide; Reference: Dulaglutide; semasita = Exposure: Semaglutide; Reference: Sitagliptin; tirzsema = Exposure: Tirzepatide; Reference: Semaglutide).

1<sup>tirzdula, semasita, tirzsema</sup> Target Trial Framework, Operational Definitions, and Data Fitness Assessment

#### 2tirzdula, semasita, tirzsema Code algorithms

2a<sup>tirzdula, semasita, tirzsema</sup> Exposure

2a<sup>tirzdula, semasita, tirzsema</sup> Inclusion

2ctirzdula, semasita, tirzsema Exclusion

2dtirzdula, semasita, tirzsema Outcome

3tirzdula, semasita, tirzsema Flowchart for cohort assembly

4tirzdula, semasita, tirzsema 1st feasibility assessment

5<sup>tirzdula, semasita, tirzsema</sup> 2nd feasibility assessment

6<sup>tirzdula, semasita, tirzsema</sup> Balance Assessment - PS Distribution and C-Statistic

 $\textbf{7}^{\text{tirzdula, semasita, tirzsema}} \, \textbf{Balance Assessment - Table 1}$ 

8<sup>tirzdula, semasita, tirzsema</sup> Covariate - Algorithm Sources

# TIRZSEMA-CVOT-SEMASITA

## **Appendices**

- 1 Target Trial Framework, Operational Definitions and Data Fitness Assessment
- 2 Code algorithms
- 2a Exposure
- 2b Inclusion
- 2c Exclusion
- 2d Outcome
- 3 Flowchart for cohort assembly
- 4 1st feasibility assessment
- 5 2nd feasibility assessment
- 6 Balance Assessment PS Distribution and C-Statistic
- 7 Balance Assessment Table 1
- 8 Covariate Algorithm Sources

| | CEMACITA | OPTUM | MADKETSCAN | MEDICARE | Notes/Overtions | Color anding |
|---|---|---|---|---|---|---|
| | SEMASITA International, double-blind, randomized, active- | Non-randomized initiation of treatment Semaglutide vs Sitagliptin | MARKETSCAN Non-randomized initiation of treatment Semaglutide vs Sitagliptin | MEDICARE Non-randomized initiation of treatment Semaglutide vs Sitagliptin | Notes/Questions | Color coding |
| index date) | controlled trial to treatment A vs B | (first eligible entry to study population) Code type: RX | (first eligible entry to study population) Code type: RX | (first eligible entry to study population) Code type: RX | | Good proxy definition |
| | | Care setting: N/A | Care setting: N/A | Care setting: N/A | | |
| | | Diagnosis position: N/A<br>Washout window: [-183,-1] | Diagnosis position: N/A<br>Washout window: [-183, -1] | Diagnosis position: N/A<br>Washout window: [-183, -1] | | |
| | | Incident with respect to: Tirzepatide in any formulation or dose Assessment window: N/A | Incident with respect to: Tirzepatide in any formulation or dose Assessment window: N/A | Incident with respect to: Tirzepatide in any formulation or dose Assessment window: N/A | | |
| | Semaglutide (subcutaneously | Source of algorithm: N/A | Source of algorithm: N/A | Source of algorithm: N/A | | |
| Exposure of | once per week) | Measurement characteristics: N/A Code type: RX | Measurement characteristics: N/A Code type: RX | Measurement characteristics: N/A<br>Code type: RX | | Moderate proxy definition |
| | | Care setting: N/A<br>Diagnosis position: N/A | Care setting: N/A<br>Diagnosis position: N/A | Care setting: N/A<br>Diagnosis position: N/A | | |
| | | Washout window: [-183, -1] | Washout window: [-183, -1] | Washout window: [-183,-1] | | |
| | | Incident with respect to: Dulaglutide in any formulation or dose Assessment window: N/A | Incident with respect to: Dulaglutide in any formulation or dose Assessment window: N/A | Incident with respect to: Dulaglutide in any formulation or dose Assessment window: N/A | | |
| Comparator 5 | Sitagliptin (oral once daily) | Source of algorithm: N/A<br>Measurement characteristics: N/A | Source of algorithm: N/A<br>Measurement characteristics: N/A | Source of algorithm: N/A<br>Measurement characteristics: N/A | | Poorly measured in database |
| · | | Code type: DX, PX | Code type: DX, PX | Code type: DX, PX | | · |
| | | Care setting: Inpatient for stroke/MI, any for death | Care setting: Inpatient for stroke/MI, any for death | Care setting: Inpatient for stroke/MI, any for death | | |
| | | Diagnosis position: Primary for Stroke, Any for MI Washout window: | Diagnosis position: Primary Washout window: | Diagnosis position: Primary for Stroke, Any for MI<br>Washout window: | | |
| | | Source of algorithm: Measurement characteristics: Death includes<br>information from the inpatient discharged dead status, social security | Source of algorithm: Measurement characteristics: Death includes information from the inpatient discharged dead status, social security | Source of algorithm: Measurement characteristics: Death includes<br>information from the inpatient discharged dead status, social security | | Poorly measured in database and not |
| Primary outcome to be emulated ! | MACE, defined as (CV death), MI, or stroke | death master file, and deaths scraped from obituaries or other sources. | death master file, and deaths scraped from obituaries or other sources. | death master file, and deaths scraped from obituaries or other sources. | | important |
| | | Code type: DX, PX Care setting: Inpatient for stroke/MI/ heart failure, any for death, | Code type: DX, PX Care setting: Inpatient for stroke/MI/ heart failure, any for death, | Code type: DX, PX Care setting: Inpatient for stroke/MI/ heart failure, any for death, | | |
| | | outpatient for i.v. diuretics Diagnosis position: Primary for stroke/ heart failure, any for MI | outpatient for i.v. diuretics Diagnosis position: Primary for stroke/ heart failure, any for MI | outpatient for i.v. diuretics Diagnosis position: Primary for stroke/ heart failure, any for MI | | |
| | | Washout window: | Washout window: | Washout window:<br>Source of algorithm: PROMISE Team, Validation studies, (Investigator | | |
| | | reviewed codes) | reviewed codes) | reviewed codes) | | |
| | | Measurement characteristics: Death includes information from the inpatient discharged dead status, social security death master file, and | Measurement characteristics: Death includes information from the inpatient discharged dead status, social security death master file, and | Measurement characteristics: Death includes information from the<br>inpatient discharged dead status, social security death master file, and | | |
| | | deaths scraped from obituaries or other sources. PPV for ischemic stroke using ICD9 codes was 88% and 95% | deaths scraped from obituaries or other sources. PPV for ischemic stroke using ICD9 codes was 88% and 95% | deaths scraped from obituaries or other sources. PPV for ischemic stroke using ICD9 codes was 88% and 95% | | |
| | | [https://pubmed.ncbi.nlm.nih.gov/12364739/ and | [https://pubmed.ncbi.nlm.nih.gov/12364739/ and | [https://pubmed.ncbi.nlm.nih.gov/12364739/ and | | |
| | | | | https://pubmed.ncbi.nlm.nih.gov/20140892/] Both of the above ICD9 codes were mapped to ICD10, but no validation | | |
| | all-cause mortality, myocardial infarction, or stroke. Composite of all-cause mortality, hospitalization for | study was performed. PPV for HHF diagnosis using ICD-10 codes was 98% in a national. | study was performed. PPV for HHF diagnosis using ICD-10 codes was 98% in a national. | study was performed. PPV for HHF diagnosis using ICD-10 codes was 98% in a national | | |
| Secondary outcome to be | | Medicare sample. | Medicare sample. | Medicare sample. | | |
| | Randomization date | One day after initiation of treatment with tirzepatide or dulaglutide | One day after initiation of treatment with tirzepatide or dulaglutide | One day after initiation of treatment with tirzepatide or dulaglutide | | |
| | | Earliest of: Outcome, end of observation in data, end of study period (365 days), discontinuation of study drug (45 days grace window and | Earliest of: Outcome, end of observation in data, end of study period (365 days), discontinuation of study drug (45 days grace window and | Earliest of: Outcome, end of observation in data, end of study period (365 days), discontinuation of study drug (45 days grace window and | | |
| Follow up end | Lyear | risk-window), switch to other GLP-1-RA, nursing home admission | risk-window), switch to other GLP-1-RA, nursing home admission | risk-window), switch to other GLP-1-RA, nursing home admission | Algorithm detail: Adherence in clinical practice databases is | |
| | | | | | expected to be much worse than in the trial, therefore the on-<br>treatment analysis at 1 year follow-up will be the primary | |
| Causal estimand | Intention-to-treat effect<br>Cox proportional hazards model | On-treatment effect Cox proportional hazards regression model | On-treatment effect Cox proportional hazards regression model | | analysis. | |
| Inclusion criteria | cox proportional nazarus model | | | | | |
| | | Applied before/after selection of index date: Before<br>Assessment window: [0, 0] | Applied before/after selection of index date: Before<br>Assessment window: [0,0] | Applied before/after selection of index date: Before<br>Assessment window: [0, 0] | | |
| | | Code type: N/A<br>Care setting: N/A | Code type: N/A<br>Care setting: N/A | Code type: N/A<br>Care setting: N/A | | |
| | | Diagnosis position: N/A<br>Source of algorithm: N/A | Diagnosis position: N/A<br>Source of algorithm: N/A | Diagnosis position: N/A<br>Source of algorithm: N/A | | |
| 1 ! | Men and women aged 18 years or older | Measurement characteristics: N/A | Measurement characteristics: N/A | Measurement characteristics: N/A | | |
| | | Applied before/after selection of index date: Before Assessment window: [-365.0] | Applied before/after selection of index date: Before Assessment window: [-365.0] | Applied before/after selection of index date: Before Assessment window: [-365.0] | | |
| | | Code type: DX<br>Care setting: Any | Code type: DX<br>Care setting: Any | Code type: DX<br>Care setting: Any | | |
| | | Diagnosis position: Any Source of algorithm: PROMISE team | Diagnosis position: Any Source of algorithm: PROMISE team | Diagnosis position: Any Source of algorithm: PROMISE team | | |
| 2 | Type 2 diabetes mellitus | Measurement characteristics: N/A | Measurement characteristics: N/A | Measurement characteristics: N/A | | |
| | | Applied before/after selection of index date: Before<br>Assessment window: [-730,0] | Applied before/after selection of index date: Before<br>Assessment window: [-730, 0] | Applied before/after selection of index date: Before<br>Assessment window: [-730,0] | | |
| | | Code type: DX, LOINC Care setting: Any | Code type: DX, LOINC Care setting: Any | Code type: DX, LOINC Care setting: Any | | |
| | | Diagnosis position: Any | Diagnosis position: Any | Diagnosis position: Any | | |
| | | Source of algorithm: Validation of obesity-related diagnosis codes in<br>claims data; Validation of body mass index (BMI)-related ICD-9-CM | Source of algorithm: Validation of obesity-related diagnosis codes in<br>claims data; Validation of body mass index (BMI)-related ICD-9-CM. | claims data; Validation of body mass index (BMI)-related ICD-9-CM | | |
| | | and ICD-10-CM administrative diagnosis codes recorded in US claims data | and ICD-10-CM administrative diagnosis codes recorded in US claims data | | Algorithm detail: If BMI measurement via LOINC code is | |
| | BMI ≥ 25kg/m2 | Measurement characteristics: N/A | Measurement characteristics: N/A | | below 10 or above 100 then measurent is set to missing. | |
| | Low, moderate, or high cardiovascular risk, definde<br>History of a cardiovascular event | | | | | |
| | | Applied before/after selection of index date: Before Assessment window: [all available data, 0] | Applied before/after selection of index date: Before Assessment window: [all available data, 0] | Applied before/after selection of index date: Before Assessment window: [all available data, 0] | | |
| | | Code type: DX | Code type: DX | Code type: DX | | |
| | | Care setting: Any<br>Diagnosis position: Any | Care setting: Any<br>Diagnosis position: Any | Care setting: Any Diagnosis position: Any | | |
| 411 | Documented history of myocardial infarction or<br>unstable angina | Source of algorithm: N/A<br>Measurement characteristics: N/A | Source of algorithm: N/A<br>Measurement characteristics: N/A | Source of algorithm: N/A<br>Measurement characteristics: N/A | | |
| 7.1.1 | | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before Assessment window: [all available data, 0] | Applied before/after selection of index date: Before Assessment window: [all available data, 0] | | |
| | | Assessment window: [all available data, 0] Code type: DX | Code type: DX | Code type: DX | | |
| | | Care setting: Any<br>Diagnosis position: Any | Care setting: Any<br>Diagnosis position: Any | Care setting: Any<br>Diagnosis position: Any | | |
| 4121 | History of ischemic stroke or TIA | Source of algorithm: N/A Measurement characteristics: N/A | Source of algorithm: N/A<br>Measurement characteristics: N/A | Source of algorithm: N/A Measurement characteristics: N/A | | |
| 4.1.2 | matory or acrieffic stroke of TIA | measurement oldi deteristics: N/A | measurement cildi deteristics; N/A | measurement cildi deteristics: IV/A | | |

| A policy of protection of the control section of related deep floride production section of related deep floride production section of related deep floride production of the control of t | | | | | |
|---|---|---|---|---|---|
| Continued of the property of | | | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before |
| Contact Cont | | | Code type: DX | | |
| Solves of injustic following and production of the control of the | | | Care setting: Any | | Care setting: Any |
| An in the comment of the anti-protects in the comment of the ant | | | Diagnosis position: Any Source of algorithm: DUPLICATE team investigator reviewed codes | Diagnosis position: Any Source of algorithm: DUPLICATE team investigator reviewed codes | Diagnosis position: Any Source of algorithm: DLIPLICATE team investigator reviewed codes |
| A Supposed my Augustian (Company of the Company of | 4.1.3 | History of heart failure | Measurement characteristics: N/A | Measurement characteristics: N/A | Measurement characteristics: N/A |
| Code types (C). If the story of project of comments on control (C) | | | | | |
| Constitution of the continue | | | | Assessment window: [all available data, 0] | |
| A second statistical processing of the second statistics of the secon | | | Care setting: Any | Care setting: Any | Care setting: Any |
| A second statistical processing of the second statistics of the secon | | | Diagnosis position: Any | Diagnosis position: Any | Diagnosis position: Any |
| Applied before wither selection or blooks date Botton Code Speec DCF, 200 Case or State Port | | | | | |
| According to an incidency of a market studency of an artification (a) Contracting or sangled file foliation of a contracting or sangled for antification (a) Contracting or sangled for antification | 4.1.4 | revascularization procedure | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before |
| Relative of control starting or singlicit Relative of control starting or singlicity | | | Assessment window: [all available data, 0] | Assessment window: [all available data, 0] | |
| Notice of control cont | | | Care setting: Any | | |
| Security of the Continue of | | | Diagnosis position: Any | Diagnosis position: Any | Diagnosis position: Any |
| Applicate before with the solution of indeed date Britished Control Section (1998) Control | | History of carotid stenting or surgical | Source of algorithm: N/A | Source of algorithm: N/A | Source of algorithm: N/A |
| Assessment without particulars of all continues and an procedure plate marked plan plant plant assessed procedure plant procedure plant plant assessed procedure plant p | 4.1.5 | revascularization | Measurement characteristics: N/A Applied before/after selection of index date: Before | Measurement characteristics: N/A Applied before/after selection of index date: Before | Measurement characteristics: N/A Applied before/after selection of index date: Before |
| The Ristory of projection was excelar procedure allowance of the Ristory of projection was excelar procedure allowance of the Ristory of projection was excellent procedure and the Ristory of projection was excellent procedure and the Ristory of projection was excellent procedure and the Ristory of projection was excellent procedure and the Ristory of projection and the Ristory of projection and the Ristory of projection and the Ristory of projection and the Ristory of projection and the Ristory of Projection and the Ristory of Carlos an | | | Assessment window: [all available data, 0] | Assessment window: [all available data, 0] | Assessment window: [all available data, 0] |
| Let be the production second production prod | | | | | |
| Selectory of procisional woundum processor designations with a contract of processor and processor | | | | | |
| Applied before order we selection or indeed date in Briton Cond-type IP. | | | Source of algorithm: N/A | Source of algorithm: N/A | Source of algorithm: N/A |
| Assessment windows pill on validation data. Q) Care setting pi N Disposis position: N/A Dis | 4.1.6 | surgical revascularization) | Measurement characteristics: N/A | Measurement characteristics: N/A | Measurement characteristics: N/A |
| Le Code type IIX. Correction of 3 antihyportensive department primary agents as defined by ACCUSANA. Applied before office of the primary agents as defined by ACCUSANA. Applied before office of the primary agents as defined by ACCUSANA. Applied before office of the primary agents as defined by ACCUSANA. Applied before office of the primary agents as defined by ACCUSANA. Assessment with deep all or validate data. Applied before office of the primary agents as defined by ACCUSANA. Assessment with deep all or validate data. Assessment with deep all or validate data. Assessment with deep all or validate data. Disposals position IVA. Disposals position IVA | | | Assessment window: [all available data 0] | Assessment window: fall available data 01 | Assessment window: [all available data 0] |
| Page 1 - 1 Documented history of contany after by discovered in particular by accordance in particular by accordan | | | Code type: RX | Code type: RX | Code type: RX |
| Source of algorithms. Printing agents as defined by ACCAMAS. Agried before other care effects. No. Measurement of survey of tables date. Before setting. No. Code type: RY. Control use of 1 in 10th ownering dring disposition of the setting. No. Code type: RY. Control use of 1 in 10th ownering dring disposition dring. Setting and the setting. No. Code type: RY. Control use of 1 in 10th ownering dring disposition dring. Setting and the setting. No. Code type: RY. Control use of 1 in 10th ownering dring disposition dring. Setting and the setting. No. Code type: RY. Control use of 1 in 10th ownering dring disposition dring. Setting and the setting. No. Code type: RY. Control use of 1 in 10th ownering dring disposition dring. Setting and the setting. No. Code type: RY. Control use of 1 in 10th ownering dring disposition dring. Setting and the setting. No. Code type: RY. Control use of 1 in 10th ownering medical and a setting. No. Code type: RY. Contr | | | | Care setting: N/A | |
| 4. Documented history of concurary arthry diseases 4. Documented history of polipheral arthry diseases 4. Documented history of polipheral arthry diseases 4. Documented history of polipheral arthry diseases 5. History of TIDM or secondary diseases 6. Receipting Arry 6. Concist years 6. Receipting Arry 6. Rece | | | Source of algorithm: Primary agents as defined by ACC/AHA | Source of algorithm: Primary agents as defined by ACC/AHA | Source of algorithm: Primary agents as defined by ACC/AHA |
| Agriel otherworks extention of fields date Biddon Accessment window; plan validate data, (1) Code type: fix Cod | | | guidelines for high blood pressure | guidelines for high blood pressure | guidelines for high blood pressure |
| Assessment window; pill available data, 0] Code to peer [N] Code to peer [ | 4.2 | Current use of ≥1 antihypertensive drug | Measurement characteristics: N/A | Measurement characteristics: N/A | Measurement characteristics: N/A |
| Code type RX Code | | | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before |
| Care settings N/A Decomposition of the story of coronary stray disease 1. Decomposition history of careful disease or disease in the stray of careful history of careful disease or disease in the stray disea | | | | | |
| Diagnosis position: N/A Source degret thera Common injudious define medications as defined and source of apport thera Common injudious define medications as defined and source of apport thera Common injudious density medications as defined and source of apport thera Common injudious density medications as defined and source of apport thera Common injudious density of the property of the selection of index date for the property of the selection of index d | | | Code type: RX | | |
| A. Durmettus of 1-tilipid kowering drug Massurement characteristics Na Massurem | | | Diagnosis position: N/A | Diagnosis position: N/A | Diagnosis position: N/A |
| Measurement tharacteristics: N/A A polleb deformation resident time. Manual production of index date Before Assessment window; plat available data, 0] Ass | | | | | |
| Applied before/after selection or findes date Before Assessment window; [all switchis data, 0] Code type; DX, C | 4.3 | Current use of ≥1 linid-lowering drug | | | |
| Learnest of the control of the contr | | our circuscor a ripid fowering drug | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before |
| A 1. Documented history of coronary artery disease A 2. Documented history of coronary artery disease A 2. Documented history of coronary artery disease A 3. Documented history of carotid artery disease A 3. Documented history of peripheral artery disease A 4. Documented history of peripheral artery disease A 4. Documented history of peripheral artery disease A 5. History of TIDM or secondary diabotes A 5. History of T | | | | | |
| A 1. Documented history of coronary artery disease A 2. Documented history of coronary artery disease A 2. Documented history of coronary artery disease A 2. Documented history of carotid artery disease A 2. Documented history of peripheral artery disease A 3. Documented history of peripheral artery disease A 3. Documented history of peripheral artery disease A 3. Documented history of peripheral artery disease A 3. Documented history of peripheral artery disease A 4. History of T1DM or secondary diabetes A 5. History of T1DM or secondary diabetes A 6. Diagnosis position. Any Diagnosis position have A 6. Diagn | | | Care setting: Any | Care setting: Any | Care setting: Any |
| Source of algorithm: N/A Documented history of coronary artery disease Applied hefore after a selection of index date Before Agriculture and a selection of index date Before Assessment window. plat available data, 0] Code type: DX Care setting: Any Source of algorithm: N/A Beginness position: Any Source of algorithm: N/A Applied hefore after a selection of index date Before Assessment window. plat available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Diagnosis | | | Diagnosis position: Any | Diagnosis position: Any | Diagnosis position: Any |
| Applied before/after selection of index date Before Assessment window [all available data, 0] Code tyne DX. Code tyne DX. Code tyne DX. Code tyne DX. Core setting: Any Source of algorithm: N/A Applied before/after selection of index date Before Assessment window [all available data, 0] Code tyne DX. Core setting: Any Source of algorithm: N/A Applied before/after selection of index date Before Assessment window. [all available data, 0] Core setting: N/A Applied before/after selection of index date Before Assessment window. [all available data, 0] Core setting: N/A Applied before/after selection of index date Before Assessment window. [all available data, 0] Core setting: Any Diagnosis position: Any Source of algorithm: N/A Applied before/after selection of index date Before Assessment window. [all available data, 0] Core setting: Any Diagnosis position: Any Source of algorithm: N/A Source of algorithm: N/A Source of algorithm: N/A Source of algorithm: N/A Measurement Anacteristics: N/A Applied before/after selection of index date Before Assessment window. [all available data, 0] Core setting: Any Diagnosis position: Any Source of algorithm: N/A Source of algorithm: N/A Measurement Anacteristics: N/A Applied before/after selection of index date Before Assessment window. [35.0] Code tyne DX Core setting: Any Source of algorithm: PGMISE team Measurement Anacteristics: N/A Applied before/after selection of index date Before Assessment window. [35.0] Code tyne DX Core setting: Any Source of algorithm: PGMISE team Measurement Anacteristics: N/A Applied before/after selection of index date Before Assessment window. [35.0] Code tyne DX Core setting: Any Diagnosis position: Any Source of algorithm: PGMISE team Measurement Anacteristics: N/A Applied before/after selection of index date Before Assessment window. [35.0] Code tyne DX, PX Core | | | Source of algorithm: N/A | Source of algorithm: N/A | Source of algorithm: N/A |
| Assessment window: [all available data, 0] Code type: DX Core setting: An Code type: DX Code ty | 4.4.1 | Documented history of coronary artery disease | | | |
| Care setting: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: N/A Applied hefore fairs selection of index date. Before | | | Assessment window: [all available data, 0] | Assessment window: [all available data, 0] | Assessment window: [all available data, 0] |
| Diagnosis position: Any Source of algorithms: N/A Source of algorithms: N/A Source of algorithms: N/A Measurement characteristics: N/A Measureme | | | Code type: DX | Code type: DX | Code type: DX |
| 4.2 Documented history of carotici artery disease Weasurement characteristics: NIA Applied before/after selection of index date: Before Assessment window: [all available data. 0] Applied before/after selection of index date: Before Assessment window: [all available data. 0] Diagnosis position: Any Source of algorithm: NIA Applied before/after selection of index date: Before Assessment window: [all available data. 0] Diagnosis position: Any Source of algorithm: NIA Measurement characteristics: NIA Applied before/after selection of index date: Before Assessment window: [all available data. 0] Diagnosis position: Any Source of algorithm: NIA Measurement characteristics: NIA Applied before/after selection of index date: Before Assessment window: [all available data. 0] Applied before/after | | | Care setting: Any Diagnosis position: Any | Diagnosis position: Any | Diagnosis position: Any |
| Applied before/after selection of index date Before Assessment window.glal valiable data, 0] Code type DX Care setting. Any Diagnosis position: Any Source of algorithms VA A3. Documented history of peripheral artery disease A4.3 Documented history of peripheral artery disease A5. Documented his | | | Source of algorithm: N/A | Source of algorithm: N/A | Source of algorithm: N/A |
| Assessment window (all available data, 0] Code type: DX Code type: DX Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Source of Algorithm: N/A Source of Algorithm: | 4.4.2 | Documented history of carotid artery disease | Measurement characteristics: N/A | Measurement characteristics: N/A | Measurement characteristics: N/A |
| Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A A.3. Documented history of peripheral artery disease Prince A.5. Documented history of peripheral artery disease Prince A.6. Survey of a position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-355, 0] Applied before/after selection of index date: Before Assessment window: [-355, 0] Assessment window: [-355, 0] Applied before/after selection of index date: Before Assessment window: [-355, 0] Assessment window: [-355, 0] Applied before/after selection of index date: Before Assessment window: [-355, 0] Code type: DX, PX Care setting: Any Diagnosis position: | | | Assessment window: [all available data: 0] | Assessment window: fall available data. 01 | Assessment window: fall available data. 01 |
| Diagnosis position: Any Source of algorithm: N/A Source of algorithm: N/A Source of algorithm: N/A Source of algorithm: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-355,0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any | | | Code type: DX | Code type: DX | Code type: DX |
| Source of algorithm: N/A Source of algorithm: N/A Measurement characteristics: N/A Measurement window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any | | | Care setting: Any | Care setting: Any | Care setting: Any |
| A.3 Documented history of peripheral artery disease Applied before/after selection of index date: Before Assessment window: [365,0] Code type: DX Care setting: Any Diagnosis position: Any Diagnosis | | | | Diagnosis position: Any Source of algorithm: N/A | Diagnosis position: Any<br>Source of algorithm: N/A |
| Applied before/after selection of index date: Before Assessment window: [-365,0] Care setting: Any Diagnosis position: Any Dia | 4.4.3 | Documented history of peripheral artery disease | | | |
| Assessment window:[-365,0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: NA Applied before/after selection of index date: Before Assessment window:[-365,0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: NA Applied before/after selection of index date: Before Assessment window:[-365,0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: NA Applied before/after selection of index date: Before Assessment window:[-365,0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement window:[-365,0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: NA Applied before/after selection of index date: Before Assessment window:[-365,0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: NA Applied before/after selection of index date: Before Assessment window:[-365,0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Applied before/after selection of index date: Before Assessment window:[-365,0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: NA Measurement characteristics: NA Applied before/after selection of index date: Before Assessment window:[-365,0] Code type: DX, PX Care setting: Any Diagnosis position: Any Diagnosis posit | teria | | Applied hefore/after selection of index data Poisson | Applied before/after selection of index data Potos | Applied before/after selection of index data: Before |
| Code type: DX Care setting: Any Diagnosis position: Any Source of algorithme PROMISE team Measurement characteristics: NA Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Source of algorithme PROMISE team Measurement characteristics: NA Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Diagnosis position | | | | | |
| Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window; [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Dia | | | Code type: DX | Code type: DX | Code type: DX |
| Surce of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Diag | | | Care setting: Any | Care setting: Any | Care setting: Any |
| S History of T10M or secondary diabetes Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: | | | Source of algorithm: PROMISE team | Source of algorithm: PROMISE team | Source of algorithm: PROMISE team |
| Assessment window: [all available data, 0] Code type: DX C | 5 | History of T1DM or secondary diabetes | Measurement characteristics: N/A | Measurement characteristics: N/A | Measurement characteristics: N/A |
| Code type: DX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Diagnosis positi | | | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before |
| Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Source of algorithm: PROMISE team Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Assessment window: [-365, | | | Code type: DX | Code type: DX | Code type: DX |
| Family or personal history of multiple endocrine 6 neoplasia or medullary thyroid carcinoma Massurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: PX Care setting: Any Diagnosis position: Any Diagnosis posi | | | Care setting: Any | Care setting: Any | Care setting: Any |
| 6 neoplasia or medullary thyroid carcinoma Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: PX Care setting: Any Diagnosis position: Any Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: PX Care setting: Any Diagnosis position: Any Measurement characteristics: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: PX Care setting: Any Diagnosis position: Any Diagnosis | | Family or personal history of acceptance | Diagnosis position: Any | Diagnosis position: Any | Diagnosis position: Any |
| Assessment window: [-365, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: PX Code type: PX Code type: PX Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Source of algorithm: PROMISE team Measurement window: [-365, 0] Code type: PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team Source of algorithm: P | | | Measurement characteristics: N/A | | |
| Code type: DX, PX Care setting: Any Diagnosis position: Any Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: PX Code type: PX Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team | | | Applied before/after selection of index date: Before | | |
| Care setting: Any Diagnosis position: Any Diagnosis po | | | | Assessment window: [-365, 0] | |
| Diagnosis position: Any Diagnosis position: Any Source of algorithme PROMISE team 7 End-stage renal disease or dialysis Measurement characteristics: N/A Measurement characteristics: N/A Measurement characteristics: N/A Measurement characteristics: N/A Measurement characteristics: N/A Applied before after selection of index date: Before Assessment window: [365.0] Assessment window: [365.0] Assessment window: [365.0] Code type: PX Code type: PX Code type: PX Code type: PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Source of algorithme PROMISE team History of treatment for diabetic retinopathy and/or Source of algorithme PROMISE team | | | Care setting: Any | Care setting: Any | Care setting: Any |
| 7 End-stagerenal disease or dialysis Measurement characteristics: N/A Measurement characteristics: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Applied before/after selection of index date: Before Assessment window: [-365,0] Applied before/after selection of index date: Before Assessment window: [-365,0] Assessment window: [-365,0] Assessment window: [-365,0] Assessment window: [-365,0] Code type: PX Code type: PX Code type: PX Code type: PX Care setting: Any Care setting: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team | | | Diagnosis position: Any | Diagnosis position: Any | Diagnosis position: Any |
| Applied before/after selection of index date: Before Assessment window: [-365,0] Code type: PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team Supplied before/after selection of index date: Before Assessment window: [-365,0] Code type: PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team Supplied before/after selection of index date: Before Assessment window: [-365,0] Code type: PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team Supplied before/after selection of index date: Before Assessment window: [-365,0] Code type: PX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team | - | End stage renal disease or dishais | Source of algorithm: PROMISE team Measurement characteristics: N/A | Source of algorithm: PROMISE team Massurament characteristics: N/A | Source of algorithm: PROMISE team |
| Assessment window: [-365,0] Assessment window: [-365,0] Assessment window: [-365,0] Code type: PX Code type: PX Code type: PX Care setting: Any Care setting: Any Care setting: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Object of algorithm: PROMISE team History of treatment for diabetic retinopathy and/or Source of algorithm: PROMISE team Source of algorithm: PROMISE team | ' | Enu-stage renar disease or dianysis | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before |
| Care setting: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team Source of algorithm: PROMISE team Source of algorithm: PROMISE team | | | Assessment window: [-365,0] | Assessment window: [-365,0] | Assessment window: [-365,0] |
| History of treatment for diabetic retinopathy and/or Source of algorithm= PROMISE team Source of algorithm= | | | | | |
| History of treatment for diabetic retinopathy and/or Source of algorithm: PROMISE team Source of algorithm: PROMISE team Source of algorithm: PROMISE team | | | Care setting: Any | | |
| 8 macular edema Measurement characteristics: N/A Measurement characteristics: N/A Measurement characteristics: N/A | | | Diagnosis position: Any | Diagnosis position: Any | Diagnosis position: Any |
| | | | Diagnosis position: Any<br>Source of algorithm: PROMISE team | Diagnosis position: Any Source of algorithm: PROMISE team | Diagnosis position: Any<br>Source of algorithm: PROMISE team |

| 9 | History of any malignancy | Applied before/after selection of Index date: Before Assessment unidow: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A | Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm PROMISE team Measurement characteristics: N/A | Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Diagnosis position: Any Obagnosis position: Any Measurement characteristics: N/A |
|---|---|---|---|---|
| 10 | Cardiovascular event or intervention in the past 7 days | | Applied before/after selection of index date: Before Assessment window: [-7, 0] Code type: DX, PX Care setting: Inpatient/ED for MI, Stroke, TIA, inpatient for procedures Diagnosis position: Any Source of algorithm: PROMISE team, Investigator reviewed codes Measurement characteristics: N/A | Applied before/after selection of index date: Before Assessment window:[-7,0] Code type: DX, PX Care setting: inpatient/ED for MI, Stroke, TIA, inpatient for procedures Diagnosis position: Any Source of algorithm: PROMISE team, investigator reviewed codes Measurement Characteristics: IN/A |
| 11 | Women who are pregnant or breastfeeding | Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A | Applied before/after selection of index date: Before Assessment windows: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A | Applied before/after selection of Index date: Before Assessment window: [-365, 0] Code type: D.X. Care setting: Arry Diagnosis position: Arry Source of algorithm: Pregnancy team Measurement Characteristics: IV/A |
| 12 | GLP-1-RA or DPP4i treatment within past 6 months | Applied before/after selection of index date: Before Assessment window: [-183, 0] Code type: RX Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: n/a | Applied before/after selection of index date: Before Assessment window: [-183, 0] Code type: RX Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: n/a | Applied before/after selection of index date: Before Assessment window: [-183, 0] Code type: RX Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: n/a |
| 13 | Bariatric surgery within the past 12 months | Applied before/after selection of index date: Before Assessment windows: [-365, 0] Code type: PX Care setting: Any Diagnosis position: Any Source of algorithms: PROMISE team Measurement character/stics: N/A | Applied before/after selection of index date: Before Assessment windows: [-365, 0] Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement character/stics: N/A | Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: P.X Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A |

Algorithm detail: Proxied by ICD-10-CM codes indicative of pregnancy at baseline.


| History of surgical or percutaneous coronary percutaneous coronary 4.14 revascularization procedure History of surgical or percutaneous coronary 4.15 revascularization procedure History of surgical or percutaneous coronary 4.16 revascularization procedure History of surgical or percutaneous coronary 4.17 revascularization procedure History of surgical or percutaneous coronary 4.18 revascularization procedure History of surgical or percutaneous coronary 4.19 revascularization procedure History of surgical or percutaneous coronary 4.10 revascularization procedure History of surgical or percutaneous coronary 4.14 revascularization procedure History of surgical or percutaneous coronary 4.15 revascularization procedure History of surgical or percutaneous coronary 4.16 revascularization procedure History of surgical or percutaneous coronary 4.17 revascularization procedure History of surgical or percutaneous coronary 4.18 revascularization procedure History of surgical or percutaneous coronary 4.19 revascularization procedure History of surgical or percutaneous coronary 4.10 revascularization procedure History of surgical or percutaneous coronary 4.14 revascularization procedure History of surgical or percutaneous coronary 4.15 revascularization procedure History of surgical or percutaneous coronary 4.16 revascularization procedure History of surgical or percutaneous coronary 4.17 revascularization procedure History of surgical or percutaneous coronary 4.18 revascularization procedure History of surgical or percutaneous coronary 4.19 revascularization procedure History of surgical or percutaneous coronary 4.10 revascularization procedure History of surgical or percutaneous coronary 4.14 revascularization procedure History of surgical or percutaneous coronary 4.15 revascularization procedure History of surgical or percutaneous coronary 4.16 revascularization procedure History of surgical or percutaneous coronary 4.17 revascularization procedure Dilla Tilon Of Coronary Artery, Two Arteries Bifurcation, Porporation of S | CD-10-PCS |
|---|---|
| 4.14 revascularization procedure History of surgical or percutaneous coronary 4.15 revascularization procedure History of surgical or percutaneous coronary 4.16 revascularization procedure History of surgical or percutaneous coronary 4.17 revascularization procedure History of surgical or percutaneous coronary 4.18 revascularization procedure History of surgical or percutaneous coronary 4.19 revascularization procedure History of surgical or percutaneous coronary 4.10 revascularization procedure History of surgical or percutaneous coronary 4.11 revascularization procedure History of surgical or percutaneous coronary 4.12 revascularization procedure History of surgical or percutaneous coronary 4.13 revascularization procedure History of surgical or percutaneous coronary 4.14 revascularization procedure History of surgical or percutaneous coronary 4.15 revascularization procedure History of surgical or percutaneous coronary 4.16 revascularization procedure History of surgical or percutaneous coronary 4.17 revascularization procedure History of surgical or percutaneous coronary 4.18 revascularization procedure History of surgical or percutaneous coronary 4.19 revascularization procedure History of surgical or percutaneous coronary 4.10 revascularization procedure History of surgical or percutaneous coronary 4.11 revascularization procedure History of surgical or percutaneous coronary 4.12 revascularization procedure History of surgical or percutaneous coronary 4.13 revascularization procedure History of surgical or percutaneous coronary 4.14 revascularization procedure History of surgical or percutaneous coronary 4.15 revascularization procedure History of surgical or percutaneous coronary 4.16 revascularization procedure History of surgical or percutaneous coronary 4.17 revascularization procedure History of surgical or percutaneous coronary 4.18 revascularization procedure History of surgical or percutaneous coronary 4.19 revascularization procedure History of surgical or percutaneous coronary 4.10 revasculariza | CD-10-PCS |
| 4.1.4 revascularization procedure History of surgical or percutaneous coronary 4.1.4 revascularization procedure Pittory of surgical or percutaneous coronary 4.1.4 revascularization procedure Pittory of surgical or percutaneous coronary 4.1.4 revascularization procedure Pittory of surgical or percutaneous coronary 4.1.4 revascularization procedure Pittory of surgical or Percutaneous coronary 4.1.4 revascularization procedure Pittory of surgical or Percutaneous c | CD-10-PCS |
| ### 4.1.4 revascularization procedure History of surgical or percutaneous coronary #### 4.1.4 revascularization procedure History of surgical or percutaneous coronary #### 4.1.4 revascularization procedure History of surgical or percutaneous coronary #### 4.1.4 revascularization | CD-10-PCS |
| 4.1.4 revascularization procedure History of surgical or percutaneous coronary 4.1.4 revascularization procedure Dilation of Coronary Artery, Two Arteries With three Drug-Ruthion of Surgical or Dilation of Coronary Artery, Two Ar | CD-10-PCS |
| Percutaneous coronary 4.1.4 revascularization procedure History of surgical or percutaneous coronary 4.1.4 revascularization procedure History of surgical or percutaneous coronary 4.1.4 revascularization procedure History of surgical or percutaneous coronary 4.1.5 revascularization procedure History of surgical or percutaneous coronary 4.1.6 revascularization procedure History of surgical or percutaneous coronary 4.1.7 revascularization procedure History of surgical or percutaneous coronary 4.1.8 revascularization procedure History of surgical or percutaneous coronary 4.1.9 revascularization procedure History of surgical or percutaneous coronary 4.1.1 revascularization procedure History of surgical or percutaneous coronary 4.1.2 revascularization procedure History of surgical or percutaneous coronary 4.1.4 revascularization procedure Parcutaneous coronary 4.1.4 revasculariza | CD-10-PCS |
| percutaneous coronary 4.1.4 revascularization procedure History of surgical or percutaneous coronary 4.1.4 revascularization procedure Picturaneous coronary 4.1.4 revascularization proce | CD-10-PCS |
| Percutaneous coronary 4.1.4 revascularization procedure History of surgical or percutaneous coronary 4.1.4 revascularization procedure Pistory of surgical or percutaneous coronary 4.1.4 revascularization procedure History of surgical or percutaneous coronary 4.1.4 revascularization procedure Pistory of surgical or percutaneous coronary 4.1.4 revascularization procedure History of surgical or percutaneous coronary 4.1.4 revascularization procedure Pistory of surgical or percutaneous coronary 4.1.4 revascularization procedure History of surgical or percutaneous coronary 4.1.4 revascularization procedure Pistory of surgical or percutaneous coronary 4.1.4 revascularization procedure History of surgical or percutaneous coronary 4.1.4 revascularization procedure History of surgical or percutaneous coronary 4.1.4 revascularization procedure Pistory of surgical or Pistory of surgi | CD-10-PCS |
| percutaneous coronary 4.1.4 revascularization procedure History of Surgical or percutaneous coronary 4.1.4 revascularization procedure D0271076 PX PX DILATION OF CORONARY ARTERY, TWO ARTERIES WITH THREE DRUG-LUTING INTRALUMINAL DEVICES, OPEN APPROACH DILATION OF CORONARY ARTERY, TWO ARTERIES, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH DILATION OF CORONARY ARTERY, TWO ARTERIES WITH FOUR OR APPROACH 4.1.4 revascularization procedure DILATION OF CORONARY ARTERY, TWO ARTERIES WITH FOUR OR APPROACH | CD-10-PCS |
| 4.1.4 revascularization procedure History of surgical or percutaneous coronary 4.1.4 revascularization procedure Dilation of Coronary Artery, Two Arteries, Bifurcation, With Four or More Drug-Eluting Intraluminal Devices, OPEN APPROACH DILATION OF CORONARY ARTERY, TWO ARTERIES, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH DILATION OF CORONARY ARTERY, TWO ARTERIES WITH FOUR OR DILATION OF CORONARY ARTERY, TWO ARTERIES WITH FOUR OR DILATION OF CORONARY ARTERY, TWO ARTERIES WITH FOUR OR DILATION OF CORONARY ARTERY, TWO ARTERIES WITH FOUR OR DILATION OF CORONARY ARTERY, TWO ARTERIES WITH FOUR OR DILATION OF CORONARY ARTERY, TWO ARTERIE | CD-10-PCS |
| 4.1.4 revascularization procedure History of surgical or percutaneous coronary 4.1.4 revascularization procedure PX APPROACH BULATION OF CORONARY ARTERY, TWO ARTERIES WITH THREE DRUG- ELUTING INTRALUMINAL DEVICES, OPEN APPROACH BULATION OF CORONARY ARTERY, TWO ARTERIES, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH BULATION OF CORONARY ARTERY, TWO ARTERIES WITH FOUR OR APPROACH BULATION OF CORONARY ARTERY, TWO ARTERIES WITH FOUR OR APPROACH BULATION OF CORONARY ARTERY, TWO ARTERIES WITH FOUR OR ALL4 revascularization procedure DILATION OF CORONARY ARTERY, TWO ARTERIES WITH FOUR OR ALL4 revascularization procedure O27107Z BULATION OF CORONARY ARTERY, TWO ARTERIES WITH FOUR OR ALL4 revascularization procedure O27107Z BULATION OF CORONARY ARTERY, TWO ARTERIES WITH FOUR OR ALL4 revascularization procedure O27107Z BULATION OF CORONARY ARTERY, TWO ARTERIES WITH FOUR OR ALL4 revascularization procedure | CD-10-PCS |
| 4.1.4 revascularization procedure History of surgical or percutaneous coronary 4.1.4 revascularization procedure Parcel | CD-10-PCS |
| 4.1.4 revascularization procedure History of surgical or percutaneous coronary 4.1.4 revascularization procedure History of surgical or percutaneous coronary 4.1.4 revascularization procedure PX History of surgical or percutaneous coronary 4.1.4 revascularization procedure PX APPROACH DILATION OF CORONARY ARTERY, TWO ARTERIES, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH DILATION OF CORONARY ARTERY, TWO ARTERIES WITH FOUR OR 4.1.4 revascularization procedure 027107Z PX MORE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH | CD-10-PCS |
| 4.1.4 revascularization procedure 0271076 PX APPROACH History of surgical or percutaneous coronary 4.1.4 revascularization procedure 027107Z PX MORE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH IN MORE DRUG-ELUTING INTRALUMINAL DEVICES DRUG-ELUTING INTR | CD-10-PCS |
| <b>4.1.4</b> revascularization procedure 027107Z PX MORE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH I | CD-10-PCS |
| History of surgical or | CD-10-PCS |
| percutaneous coronary DILATION OF CORONARY ARTERY, TWO ARTERIES, BIFURCATION, | CD-10-PCS |
| percutaneous coronary DILATION OF CORONARY ARTERY, TWO ARTERIES WITH | CD-10-PCS |
| percutaneous coronary DILATION OF CORONARY ARTERY, TWO ARTERIES, BIFURCATION, | CD-10-PCS |


| | | | TRANSCATHETER PLACEMENT OF AN INTRACO | DONA DV STENT/S) |
|---|---|---|---|---|
| History of surgical or | | | PERCUTANEOUS, WITH OR WITHOUT OTHER THE | |
| percutaneous coronary | / | | INTERVENTION, ANY METHOD; EACH ADDITIONA | |
| <b>4.1.4</b> revascularization proce | | 92981 P | SEPARATELY IN ADDITION TO CODE FOR PRIMAR | • |
| History of surgical or | | | | , |
| percutaneous coronary | / | | PERCUTANEOUS TRANSLUMINAL CORONARY B. | ALLOON |
| <b>4.1.4</b> revascularization proce | edure | 92982 P | ANGIOPLASTY; SINGLE VESSEL | ICD-10-PCS |
| History of surgical or | | | PERCUTANEOUS TRANSLUMINAL CORONARY B. | ALLOON |
| percutaneous coronary | | | ANGIOPLASTY; EACH ADDITIONAL VESSEL (LIST | |
| 4.1.4 revascularization proce | edure | 92984 P | ADDITION TO CODE FOR PRIMARY PROCEDURE) | |
| History of surgical or | | | PERCUTANEOUS TRANSLUMINAL CORONARY A | |
| percutaneous coronary | | | MECHANICAL OR OTHER METHOD, WITH OR WITH | |
| 4.1.4 revascularization proce | edure | 92995 P | ANGIOPLASTY; SINGLE VESSEL | ICD-10-PCS |
| Historyoformaladay | | | PERCUTANEOUS TRANSLUMINAL CORONARY A | |
| History of surgical or | | | MECHANICAL OR OTHER METHOD, WITH OR WITH | |
| percutaneous coronary <b>4.1.4</b> revascularization proce | | 92996 P | ANGIOPLASTY; EACH ADDITIONAL VESSEL (LIST<br>ADDITION TO CODE FOR PRIMARY PROCEDURE) | |
| History of surgical or | edule | 32330 F | ADDITION TO CODE FOR FRIMART FROCEDORE) | ICD-10-F C3 |
| percutaneous coronary | / | | | |
| <b>4.1.4</b> revascularization proce | | D) | PRESENCE OF AORTOCORONARY BYPASS GRAF | T ICD-10-PCS |
| History of surgical or | | | | |
| percutaneous coronary | / | | | |
| 4.1.4 revascularization proce | edure Z95.5 | D) | PRESENCE OF CORONARY ANGIOPLASTY IMPLA | ANT AND GRAFT ICD-10-PCS |
| History of surgical or | | | | |
| percutaneous coronary | | | | |
| 4.1.4 revascularization proce | | 1 D | CORONARY ANGIOPLASTY STATUS | ICD-10-PCS |
| History of carotid sten | _ | | BYPASS RIGHT COMMON CAROTID ARTERY TO IT | |
| 4.1.5 surgical revascularizat | | 09G P | ARTERY WITH AUTOLOGOUS VENOUS TISSUE, OF | |
| History of carotid sten | | ) A C D) | BYPASS RIGHT COMMON CAROTID ARTERY TO IT | |
| 4.1.5 surgical revascularizat<br>History of carotid sten | | DAG P | ARTERY WITH AUTOLOGOUS ARTERIAL TISSUE,<br>BYPASS RIGHT COMMON CAROTID ARTERY TO I | |
| 4.1.5 surgical revascularizat | | OJG P | ARTERY WITH SYNTHETIC SUBSTITUTE, OPEN AF | |
| 4.1.3 Suigicai revascularizat | 051110 | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | BYPASS RIGHT COMMON CAROTID ARTERY TO IT | |
| History of carotid sten | ting or | | ARTERY WITH NONAUTOLOGOUS TISSUE SUBST | |
| 4.1.5 surgical revascularizat | | OKG P | APPROACH | ICD-10-PCS |
| History of carotid sten | ting or | | BYPASS RIGHT COMMON CAROTID ARTERY TO IT | NTRACRANIAL |
| 4.1.5 surgical revascularizat | ion 031HC | DZG PX | ARTERY, OPEN APPROACH | ICD-10-PCS |
| History of carotid sten | _ | | BYPASS LEFT COMMON CAROTID ARTERY TO IN | |
| 4.1.5 surgical revascularizat | | 9G P | ARTERY WITH AUTOLOGOUS VENOUS TISSUE, OF | |
| History of carotid sten | _ | | BYPASS LEFT COMMON CAROTID ARTERY TO IN | |
| 4.1.5 surgical revascularizat | | AG P | ARTERY WITH AUTOLOGOUS ARTERIAL TISSUE, | |
| History of carotid sten | | JG P | BYPASS LEFT COMMON CAROTID ARTERY TO IN | |
| 4.1.5 surgical revascularizat | 1011 03110 | JG P | ARTERY WITH SYNTHETIC SUBSTITUTE, OPEN AF<br>BYPASS LEFT COMMON CAROTID ARTERY TO IN | |
| History of carotid sten | ting or | | ARTERY WITH NONAUTOLOGOUS TISSUE SUBST | |
| 4.1.5 surgical revascularizat | | KG P | APPROACH | ICD-10-PCS |
| History of carotid stem | | | BYPASS LEFT COMMON CAROTID ARTERY TO IN | |
| 4.1.5 surgical revascularizat | | ZG P | ARTERY, OPEN APPROACH | ICD-10-PCS |
| History of carotid sten | | | DILATION OF INTRACRANIAL ARTERY WITH DRU | G-ELUTING |
| 4.1.5 surgical revascularizat | ion 037G0 | 04Z P | INTRALUMINAL DEVICE, OPEN APPROACH | ICD-10-PCS |
| History of carotid sten | ting or | | DILATION OF INTRACRANIAL ARTERY WITH TWO | |
| 4.1.5 surgical revascularizat | | 05Z P | INTRALUMINAL DEVICE, OPEN APPROACH | ICD-10-PCS |
| History of carotid sten | | | DILATION OF INTRACRANIAL ARTERY WITH THR | |
| 4.1.5 surgical revascularizat | | 06Z P | INTRALUMINAL DEVICE, OPEN APPROACH | ICD-10-PCS |
| History of carotid sten | _ | 077 | DILATION OF INTRACRANIAL ARTERY WITH FOU | |
| 4.1.5 surgical revascularizat | | 07Z P | ELUTING INTRALUMINAL DEVICE, OPEN APPROA | |
| History of carotid sten 4.1.5 surgical revascularizat | | ODZ P | DILATION OF INTRACRANIAL ARTERY WITH INTR<br>OPEN APPROACH | RALUMINAL DEVICE, ICD-10-PCS |
| T.I.J Surgical revascularizat | 1011 03/60 | UDZ P | UPENAFRUACH | ICD-10-PC3 |


| History of peripheral vascular procedure (sterling or surgical Mistory of peripheral vascular | | | | | | |
|---|---|---|---|---|---|---|
| 4.16 revascularization) Octobrol vascular procedure (sterning or surgical 4.16 revascularization) History of peripheral vascular pro | | History of peripheral vascular | | | | |
| 4.16 revascularization) Octobrol vascular procedure (sterning or surgical 4.16 revascularization) History of peripheral vascular pro | | procedure (stenting or surgical | | | EXTIRPATION OF MATTER FROM RIGHT POPLITEAL ARTERY, OPEN | |
| History of peripheral vascular procedure (sterning or sugical | 4.1.6 | | 04CM0ZZ | PX | | ICD-10-PCS |
| procedure (steming or sugical 4.16 revascularization) History of peripheral vascular proced | | | | | | |
| ## STIRPATION OF MATTER FROM LEFT POPLITEAL ARTERY, DPS DEFUNCATION, PERCUTANEOUS APPROACH (ICD-10-PCS History of peripheral vascular procedure (sterning or surgical AL16 revascularization) | | | | | EXTIREATION OF MATTER FROM RIGHT POPI ITEAL ARTERY | |
| History of peripheral vascular procedure festering or surgical History of peripheral vascular procedure festering or surgical History of peripheral vascular procedure festering or surgical A1.6 revascularization) 41.6 revascularization O4CM4Z6 PX BIFURCATION OF MATTER FROM RIGHT POPLITEAL ARTERY, PERCUTANEOUS ENDOSCOPIC APPROACH ICD-10-PCS HISTORY OF peripheral vascular procedure festering or surgical Procedure festering or surgical Procedure festering or surgical Procedure festering or surgical History of peripheral vascular procedure festering or surgical Procedure festering or surgical Procedure festering or surgical Procedure festering or surgical Procedure festering or surgical Procedure festering or surgical History of peripheral vascular procedure festering or surgical Procedure festering or surgical | 410 | | 0.4014270 | DV | | ICD 10 DCC |
| Procedure istenting or surgical 4.16 revascularization) History of peripheral vascular procedure (stenting or surgical 4.16 revascul | 4.1.6 | | 04CM3Z6 | PX | BIFURCATION, PERCUTANEOUS APPROACH | ICD-10-PCS |
| 4.16 revascularization) Oct Max 2 PX PERCUTANEOUS APPROACH (ICD-10-PCS History of peripheral vascular procedure (stenting or surgical 4.16 revascularization) History of peripheral vascular procedure (stenting or surgical 4.16 revascularization) Peripheral vascular Peripheral vascular procedure (stenting or surgical 4.16 revascularization) Peripheral vascular Peripheral va | | | | | EVERDATION OF MATTER EDOMARIOUT DODLUTEM ADTERV | |
| History of peripheral vascular procedure festering or surgical History of peripheral vascular | | | | | | |
| procedure(sterting or surgical 4.16. revascularization) History of peripheral vascular procedure(sterting or surgical 4.16. revascul | 4.1.6 | • | 04CM3ZZ | PX | PERCUTANEOUS APPROACH | ICD-10-PCS |
| 4.1.6 revascularization) deCM4Z6 PX BIFURCATION_PERCUTANEOUS ENDOSCOPIC APPROACH (CD-10-PCS PROCEDURE) PROCEDURE (Sterting or surgical AL.6 revascularization) History of peripheral vascular procedure (sterting or surgical AL.6 revascularization) History of peripheral vascular procedure (sterting or surgical AL.6 revascularization) History of peripheral vascular procedure (sterting or surgical AL.6 revascularization) History of peripheral vascular procedure (sterting or surgical AL.6 revascularization) History of peripheral vascular procedure (sterting or surgical History of peripheral vascular procedure (sterting or surgical AL.6 revascularization) History of peripheral vascular procedure (sterting or surgical His | | | | | | |
| 4.1.6 revascularization) deCM4Z6 PX BIFURCATION_PERCUTANEOUS ENDOSCOPIC APPROACH (CD-10-PCS PROCEDURE) PROCEDURE (Sterting or surgical AL.6 revascularization) History of peripheral vascular procedure (sterting or surgical AL.6 revascularization) History of peripheral vascular procedure (sterting or surgical AL.6 revascularization) History of peripheral vascular procedure (sterting or surgical AL.6 revascularization) History of peripheral vascular procedure (sterting or surgical AL.6 revascularization) History of peripheral vascular procedure (sterting or surgical History of peripheral vascular procedure (sterting or surgical AL.6 revascularization) History of peripheral vascular procedure (sterting or surgical His | | procedure (stenting or surgical | | | EXTIRPATION OF MATTER FROM RIGHT POPLITEAL ARTERY, | |
| History of peripheral vascular procedure (stenting or surgical 4.1.6 revascular/zation) | 4.1.6 | | 04CM4Z6 | PX | BIFURCATION. PERCUTANEOUS ENDOSCOPIC APPROACH | ICD-10-PCS |
| procedure (stenting or surgical 4.1.6 revascularization) History of peripheral vascular procedure (stenting or | | History of peripheral vascular | | | | |
| ### ACCUPATION OF MATTER FROM LEFT POPLITEAL ARTERY, OPEN BIFURCATION, OPEN APPROACH ### APPROACH | | | | | EXTIRPATION OF MATTER FROM RIGHT POPLITEAL ARTERY | |
| History of peripheral vascular procedure (sterning or surgical | 116 | | 040M477 | DV | | ICD 10 DCS |
| procedure (sterning or surgical 4.16. revascularization) History of peripheral vascular procedure (sterning or | 4.1.0 | • | U4CIVI4ZZ | FX | PENCOTANLOUS ENDOSCOPIC APPROACIT | ICD-10-F C3 |
| ### ALIA revascularization History of peripheral vascular procedure (sterting or surgical His | | | | | EVERDATION OF MATTER EDOM SET DOD UTEM ADTERV | |
| History of peripheral vascular procedure (stertling or surgical pr | | | | | · | |
| ### STIRPATION OF MATTER FROM LEFT POPLITEAL ARTERY, OPEN ### APPROACH STIRPATION OF MATTER FROM LEFT POPLITEAL ARTERY, OPEN ### APPROACH STIRPATION OF MATTER FROM LEFT POPLITEAL ARTERY, OPEN ### APPROACH STIRPATION OF MATTER FROM LEFT POPLITEAL ARTERY, OPEN ### APPROACH STIRPATION OF MATTER FROM LEFT POPLITEAL ARTERY, OPEN ### APPROACH STIRPATION OF MATTER FROM LEFT POPLITEAL ARTERY, OPEN ### ALIGN or versus clarization OACN3ZZ PX PERCUTANEOUS APPROACH ICD-10-PCS ### History of peripheral vascular procedure (stenting or surgical Procedure (stenting | 4.1.6 | • | 04CN0Z6 | PX | BIFURCATION, OPEN APPROACH | ICD-10-PCS |
| 4.1.6 revascularization) | | History of peripheral vascular | | | | |
| History of peripheral vascular procedure (stenting or surgical History of peripheral vascular procedure (stenting or surgical History of peripheral vascular procedure (stenting or surgical History of peripheral vascular procedure (stenting or surgical History of peripheral vascular procedure (stenting or surgical Procedure (stenting or surgical Pro | | procedure (stenting or surgical | | | EXTIRPATION OF MATTER FROM LEFT POPLITEAL ARTERY, OPEN | |
| 4.16 revascularization) 4.17 revascularization) 4.18 revascularization) 4.19 revascularization) 4.10 revascularization) 4.10 revascularization) 4.10 revascularization) 4.11 revascularization) 4.12 revascularization) 4.13 revascularization) 4.14 revascularization) 4.15 revascularization) 4.16 revascularization) 4.16 revascularization) 4.17 revascularization) 4.18 revascularization) 4.19 revascularization) 4.10 revascularization) 4.10 revascularization) 4.10 revascularization) 4.11 revascularization) 4.12 revascularization) 4.13 revascularization) 4.14 revascularization) 4.15 revascularization) 4.16 revascularization) 4.17 revascularization) 4.18 revascularization) 4.19 revascularization) 4.19 revascularization) 4.10 revascularization) 4.10 revascularization) 4.11 revascularization) 4.12 revascularization) 4.13 revascularization) 4.14 revascularization) 4.15 revascularization) 4.16 revascularization) 4.17 revascularization) 4.18 revascularization) 4.19 revascularization) 4.19 revascularization) 4.10 revascularization) 4.11 revascularization) 4.12 revascularization) 4.13 revascularization) 4.14 revascularization) 4.15 revascularization) 4.16 revascularization) 4.17 revascularization) 4.18 revascularization) 4.19 revascularization) 4.19 revascularization) 4.10 revascularization) 4.11 revascularization) 4.12 revascularization) 4.13 revascularization) 4.14 revascularization) 4.15 revascularization) 4.16 revascularization) 4.17 revascularization) 4.18 revascularization) 4.19 revascularization) 4.19 revascularization) 4.10 revascularization) 4.11 revascularization) 4.12 revascularization) 4.13 revascularization) 4.14 r | 4.1.6 | revascularization) | 04CN0ZZ | PX | APPROACH | ICD-10-PCS |
| 4.16 revascularization) 4.17 revascularization) 4.18 revascularization) 4.19 revascularization) 4.10 revascularization) 4.10 revascularization) 4.10 revascularization) 4.11 revascularization) 4.12 revascularization) 4.13 revascularization) 4.14 revascularization) 4.15 revascularization) 4.16 revascularization) 4.16 revascularization) 4.17 revascularization) 4.18 revascularization) 4.19 revascularization) 4.10 revascularization) 4.10 revascularization) 4.10 revascularization) 4.11 revascularization) 4.12 revascularization) 4.13 revascularization) 4.14 revascularization) 4.15 revascularization) 4.16 revascularization) 4.17 revascularization) 4.18 revascularization) 4.19 revascularization) 4.19 revascularization) 4.10 revascularization) 4.10 revascularization) 4.11 revascularization) 4.12 revascularization) 4.13 revascularization) 4.14 revascularization) 4.15 revascularization) 4.16 revascularization) 4.17 revascularization) 4.18 revascularization) 4.19 revascularization) 4.19 revascularization) 4.10 revascularization) 4.11 revascularization) 4.12 revascularization) 4.13 revascularization) 4.14 revascularization) 4.15 revascularization) 4.16 revascularization) 4.17 revascularization) 4.18 revascularization) 4.19 revascularization) 4.19 revascularization) 4.10 revascularization) 4.11 revascularization) 4.12 revascularization) 4.13 revascularization) 4.14 revascularization) 4.15 revascularization) 4.16 revascularization) 4.17 revascularization) 4.18 revascularization) 4.19 revascularization) 4.19 revascularization) 4.10 revascularization) 4.11 revascularization) 4.12 revascularization) 4.13 revascularization) 4.14 r | | History of peripheral vascular | | | | |
| ### ACC 10-10-PCS History of peripheral vascular procedure (stenting or surgical History of peripheral vascular procedure (stenting or surgical Procedure (ste | | | | | EXTIRPATION OF MATTER FROM LEFT POPLITEAL ARTERY | |
| History of peripheral vascular procedure (stenting or surgical A1.6 revascularization) History of peripheral vascular procedure (stenting or surgical History of peripheral vascular procedure (stenting or surgical Pistory of peripheral vascular procedure (stenting or surgical History of peripheral vascular procedure (stenting or surgical Procedure (stentin | 416 | | 0400376 | DY | · | ICD-10-PCS |
| ### A1.6 revascularization ### A1.6 revasculariz | 4.1.0 | | 04011320 | 1 % | BII DICATION, I EICOTANEOUS AIT IOACH | ICD-10-1 C3 |
| History of peripheral vascular procedure (stenting or surgical A1.6 revascularization) History of peripheral vascular procedure (stenting or surgical Procedure (stenting or surgical Procedur | | | | | EVIDDATION OF MATTER EDOM LEFT DODL ITEM. ADTERV | |
| History of peripheral vascular procedure (stenting or surgical A.1.6 revascularization) History of peripheral vascular procedure (stenting or surgical Procedure (stenting or surgical Procedu | | | | 5.4 | | 100 40 000 |
| ### A1.6 revascularization of peripheral vascular procedure (stenting or surgical History of peripheral vascular procedure (stenting or surgical History of peripheral vascular procedure (stenting or surgical Procedure (ste | 4.1.6 | • | U4CN3ZZ | PX | PERCUTANEOUS APPROACH | ICD-10-PCS |
| ### A1.6 revascularization | | | | | | |
| History of peripheral vascular procedure (stenting or surgical History of peripheral vascular procedure (stenting or surgical History of peripheral vascular procedure (stenting or surgical History of peripheral vascular procedure (stenting or surgical Procedure (stenting or surgical History of peripheral vascular procedure (stenting or surgical Procedure (stenting or surgical History of peripheral vascular procedure (stenting or surgical Procedure (stenting or surgical Proc | | | | | | |
| ## A.1.6 revascularization ## A.1.6 revascularization ## A.1.6 revascularization ## A.1.6 revascularization ## PERCUTANEOUS ENDOSCOPIC APPROACH ## ISTORY of peripheral vascular ## procedure (stenting or surgical ## A.1.6 revascularization ## A.1.6 revascularization ## PERCUTANEOUS ENDOSCOPIC APPROACH ## ISTORY OF peripheral vascular ## procedure (stenting or surgical ## A.1.6 revascularization ## PERCUTANEOUS ENDOSCOPIC APPROACH ## ISTORY OF peripheral vascular ## procedure (stenting or surgical ## A.1.6 revascularization ## A.1.6 revascularization ## A.1.6 revascularization ## PERCUTANEOUS APPROACH ## ISTORY OF PERCUTANEOUS ENDOSCOPIC APPROACH ## ISTORY OF PERCUTANEOUS E | 4.1.6 | revascularization) | 04CN4Z6 | PX | BIFURCATION, PERCUTANEOUS ENDOSCOPIC APPROACH | ICD-10-PCS |
| 4.1.6 revascularization) 04CN4ZZ PX PERCUTANEOUS ENDOSCOPIC APPROACH ICD-10-PCS History of peripheral vascular procedure (stenting or surgical stenting or surgical procedure (stenting or surgical stenting | | History of peripheral vascular | | | | |
| 4.1.6 revascularization) 04CN4ZZ PX PERCUTANEOUS ENDOSCOPIC APPROACH ICD-10-PCS History of peripheral vascular procedure (stenting or surgical stenting or surgical procedure (stenting or surgical stenting | | procedure (stenting or surgical | | | EXTIRPATION OF MATTER FROM LEFT POPLITEAL ARTERY. | |
| History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) History of peripheral vascular procedure (stenting or surgical procedure (stenting or surgical 4.1.6 revascularization) History of peripheral vascular procedure (stenting or surgical procedure (stenting or surgical 4.1.6 revascularization) History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) O4CP3ZZ PX History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) O4CP3ZZ PX History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) O4CP4ZE PX History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) O4CP4ZE PX History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) O4CP4ZE PX History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) O4CP4ZZ PX History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) O4CP4ZZ PX PX PERCUTANEOUS ENDOSCOPIC APPROACH ICD-10-PCS History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) O4CP4ZZ PX PERCUTANEOUS ENDOSCOPIC APPROACH ICD-10-PCS History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) O4CP4ZZ PX PERCUTANEOUS ENDOSCOPIC APPROACH ICD-10-PCS History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) O4CP4ZZ PX PERCUTANEOUS ENDOSCOPIC APPROACH ICD-10-PCS History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) O4CP4ZZ PX PERCUTANEOUS ENDOSCOPIC APPROACH ICD-10-PCS BIFURCATION, OPEN APPROACH ICD-10-PCS BIFURCATION, OPEN APPROACH ICD-10-PCS BIFURCATION, OPEN APPROACH ICD-10-PCS BIFURCATI | 4.1.6 | | 04CN4ZZ | PX | PERCUTANEOUS ENDOSCOPIC APPROACH | ICD-10-PCS |
| 4.1.6 revascularization) O4CPOZE PX BIFURCATION OF MATTER FROM RIGHT ANTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH ICD-10-PCS History of peripheral vascular procedure (stenting or surgical procedure (stenting or surgi | | | | | | |
| 4.1.6 revascularization) 04CP0Z6 PX BIFURCATION, OPEN APPROACH ICD-10-PCS History of peripheral vascular procedure (stenting or surgical procedure (stenting o | | | | | EXTIREATION OF MATTER FROM RIGHT ANTERIOR TIRIAL ARTERY | |
| History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) History of peripheral vascular procedure (stenting or surgical procedure (stenting or surgical 4.1.6 revascularization) History of peripheral vascular procedure (stenting or surgical procedure (stenting or surgical 4.1.6 revascularization) 4.1.6 revascularization) History of peripheral vascular procedure (stenting or surgical standard procedure (stenting or surgical procedure (stenting or surgical standard procedure (stentin | 416 | | 0.400.76 | DV | · · | ICD 10 DCC |
| ### A1.6 revascularization of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) | 4.1.6 | | U4CPUZ6 | PX | BIFURCATION, OPEN APPROACH | ICD-10-PCS |
| 4.1.6 revascularization) 04CP0ZZ PX OPENAPPROACH ICD-10-PCS History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) 04CP3Z6 PX BIFURCATION OF MATTER FROM RIGHT ANTERIOR TIBIAL ARTERY, History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) 04CP3Z2 PX PERCUTANEOUS APPROACH ICD-10-PCS History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) 04CP4Z6 PX BIFURCATION OF MATTER FROM RIGHT ANTERIOR TIBIAL ARTERY, History of peripheral vascular procedure (stenting or surgical procedure (stenting or surgical 4.1.6 revascularization) 04CP4Z6 PX BIFURCATION OF MATTER FROM RIGHT ANTERIOR TIBIAL ARTERY, History of peripheral vascular procedure (stenting or surgical procedure (stenting or surgical 4.1.6 revascularization) 04CP4Z2 PX PERCUTANEOUS ENDOSCOPIC APPROACH ICD-10-PCS History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) 04CP4Z6 PX PERCUTANEOUS ENDOSCOPIC APPROACH ICD-10-PCS EXTIRPATION OF MATTER FROM LEFT ANTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH ICD-10-PCS EXTIRPATION OF MATTER FROM LEFT ANTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH ICD-10-PCS EXTIRPATION OF MATTER FROM LEFT ANTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH ICD-10-PCS EXTIRPATION OF MATTER FROM LEFT ANTERIOR TIBIAL ARTERY, EXTIRPATION OF MATTER FROM LEFT ANTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH ICD-10-PCS EXTIRPATION OF MATTER FROM LEFT ANTERIOR TIBIAL ARTERY, EXTIRPATION OF MATTER FROM LEFT ANTERIOR TIB | | | | | EVERDATION OF MATTER EDOMARIANT ANTERIOR TIDIAL ARTERY | |
| History of peripheral vascular procedure (stenting or surgical revascularization) | | | | | | |
| ### Procedure (stenting or surgical 4.1.6 revascularization) | 4.1.6 | • | 04CP0ZZ | PX | OPEN APPROACH | ICD-10-PCS |
| 4.1.6 revascularization) 04CP3Z6 PX BIFURCATION, PERCUTANEOUS APPROACH ICD-10-PCS History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) 04CP3ZZ PX PERCUTANEOUS APPROACH ICD-10-PCS History of peripheral vascular procedure (stenting or surgical procedure | | History of peripheral vascular | | | | |
| History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) | | procedure (stenting or surgical | | | EXTIRPATION OF MATTER FROM RIGHT ANTERIOR TIBIAL ARTERY, | |
| History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) | 4.1.6 | revascularization) | 04CP3Z6 | PX | BIFURCATION, PERCUTANEOUS APPROACH | ICD-10-PCS |
| procedure (stenting or surgical revascularization) | | | | | | |
| 4.1.6 revascularization) 04CP3ZZ PX PERCUTANEOUS APPROACH ICD-10-PCS History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) 04CP4Z6 PX BIFURCATION OF MATTER FROM RIGHT ANTERIOR TIBIAL ARTERY, History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) 04CP4Z2 PX PERCUTANEOUS ENDOSCOPIC APPROACH ICD-10-PCS History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) 04CP4ZZ PX PERCUTANEOUS ENDOSCOPIC APPROACH ICD-10-PCS History of peripheral vascular procedure (stenting or surgical EXTIRPATION OF MATTER FROM LEFT ANTERIOR TIBIAL ARTERY, History of peripheral vascular procedure (stenting or surgical EXTIRPATION OF MATTER FROM LEFT ANTERIOR TIBIAL ARTERY, History of peripheral vascular procedure (stenting or surgical EXTIRPATION OF MATTER FROM LEFT ANTERIOR TIBIAL ARTERY, | | | | | EXTIRPATION OF MATTER FROM RIGHT ANTERIOR TIRIAL ARTERY | |
| History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) 04CP4Z6 PX BIFURCATION OF MATTER FROM RIGHT ANTERIOR TIBIAL ARTERY, History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) 04CP4ZZ PX PERCUTANEOUS ENDOSCOPIC APPROACH ICD-10-PCS History of peripheral vascular procedure (stenting or surgical Procedure (stenting | 416 | | 04CP377 | PX | | ICD-10-PCS |
| procedure (stenting or surgical revascularization) 04CP4Z6 PX BIFURCATION OF MATTER FROM RIGHT ANTERIOR TIBIAL ARTERY, History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) 04CP4ZZ PX PERCUTANEOUS ENDOSCOPIC APPROACH ICD-10-PCS History of peripheral vascular procedure (stenting or surgical Procedure (stenting or su | 7.1.0 | • | 0 101 JLL | 1.7 | 1 ENGO MILEGOOM I NOMON | 100 10 1 00 |
| 4.1.6 revascularization) 04CP4Z6 PX BIFURCATION, PERCUTANEOUS ENDOSCOPIC APPROACH ICD-10-PCS History of peripheral vascular procedure (stenting or surgical EXTIRPATION OF MATTER FROM RIGHT ANTERIOR TIBIAL ARTERY, 4.1.6 revascularization) 04CP4ZZ PX PX PERCUTANEOUS ENDOSCOPIC APPROACH ICD-10-PCS History of peripheral vascular procedure (stenting or surgical EXTIRPATION OF MATTER FROM LEFT ANTERIOR TIBIAL ARTERY, ICD-10-PCS History of peripheral vascular procedure (stenting or surgical PX BIFURCATION, OPEN APPROACH ICD-10-PCS EXTIRPATION OF MATTER FROM LEFT ANTERIOR TIBIAL ARTERY, EXTIRPATION OF MATTER FROM LEFT ANTERIOR TIBIAL ARTERY, ICD-10-PCS | | | | | EVTIDDATION OF MATTED FROM BIOLIT ANTERIOR TIDIAL ARTERY | |
| History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) 04CP4ZZ PX PERCUTANEOUS ENDOSCOPIC APPROACH ICD-10-PCS History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) 04CQ0Z6 PX BIFURCATION, OPEN APPROACH ICD-10-PCS BIFURCATION ICD-10-PCS BIFUR | | | 0.400.476 | DV | · · | 100 10 000 |
| procedure (stenting or surgical 4.1.6 revascularization) 04CP4ZZ PX PERCUTANEOUS ENDOSCOPIC APPROACH ICD-10-PCS History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) 04CQ0Z6 PX BIFURCATION OF MATTER FROM LEFT ANTERIOR TIBIAL ARTERY, History of peripheral vascular procedure (stenting or surgical EXTIRPATION OF MATTER FROM LEFT ANTERIOR TIBIAL ARTERY, EXTIRPATION OF MATTER FROM LEFT ANTERIOR TIBIAL ARTERY, EXTIRPATION OF MATTER FROM LEFT ANTERIOR TIBIAL ARTERY, EXTIRPATION OF MATTER FROM LEFT ANTERIOR TIBIAL ARTERY, EXTIRPATION OF MATTER FROM LEFT ANTERIOR TIBIAL ARTERY, | 4.1.6 | | 04CP4Z6 | PX | BIFURCATION, PERCUTANEOUS ENDOSCOPIC APPROACH | ICD-10-PCS |
| 4.1.6 revascularization) 04CP4ZZ PX PERCUTANEOUS ENDOSCOPIC APPROACH ICD-10-PCS History of peripheral vascular procedure (stenting or surgical) 4.1.6 revascularization) 04CQ0Z6 PX BIFURCATION, OPEN APPROACH ICD-10-PCS History of peripheral vascular procedure (stenting or surgical) EXTIRPATION OF MATTER FROM LEFT ANTERIOR TIBIAL ARTERY, ICD-10-PCS | | | | | | |
| History of peripheral vascular procedure (stenting or surgical EXTIRPATION OF MATTER FROM LEFT ANTERIOR TIBIAL ARTERY, 4.1.6 revascularization) 04CQ0Z6 PX BIFURCATION, OPEN APPROACH ICD-10-PCS History of peripheral vascular procedure (stenting or surgical EXTIRPATION OF MATTER FROM LEFT ANTERIOR TIBIAL ARTERY, | | | | | | |
| procedure (stenting or surgical 4.1.6 revascularization) 04CQ0Z6 PX BIFURCATION, OPEN APPROACH ICD-10-PCS History of peripheral vascular procedure (stenting or surgical EXTIRPATION OF MATTER FROM LEFT ANTERIOR TIBIAL ARTERY, EXTIRPATION OF MATTER FROM LEFT ANTERIOR TIBIAL ARTERY, | 4.1.6 | revascularization) | 04CP4ZZ | PX | PERCUTANEOUS ENDOSCOPIC APPROACH | ICD-10-PCS |
| procedure (stenting or surgical 4.1.6 revascularization) 04CQ0Z6 PX BIFURCATION, OPEN APPROACH ICD-10-PCS History of peripheral vascular procedure (stenting or surgical EXTIRPATION OF MATTER FROM LEFT ANTERIOR TIBIAL ARTERY, EXTIRPATION OF MATTER FROM LEFT ANTERIOR TIBIAL ARTERY, | | History of peripheral vascular | | | | |
| 4.1.6 revascularization) 04CQ0Z6 PX BIFURCATION, OPEN APPROACH ICD-10-PCS History of peripheral vascular procedure (stenting or surgical EXTIRPATION OF MATTER FROM LEFT ANTERIOR TIBIAL ARTERY, | | | | | EXTIRPATION OF MATTER FROM LEFT ANTERIOR TIBIAL ARTERY. | |
| History of peripheral vascular procedure (stenting or surgical EXTIRPATION OF MATTER FROM LEFT ANTERIOR TIBIAL ARTERY, | 4.1.6 | | 04C00Z6 | PX | | ICD-10-PCS |
| procedure (stenting or surgical EXTIRPATION OF MATTER FROM LEFT ANTERIOR TIBIAL ARTERY, | | | 04020 | | | 10 . 00 |
| | | | | | EYTIRDATION OF MATTER FROM LEFT ANTERIOR TIDIAL ADTEDV | |
| T.I.O TEVASCULARIZATION U4CQUZZ FA OPENAPPROACH ICD-10-PCS | 410 | | 0400077 | DV | | ICD 10 DCC |
| | 4.1.0 | revascularizationij | UHCQUZZ | ΓΛ | OF LIVAF FIVOACH | ICD-10-LC2 |


REVASCULARIZATION, ENDOVASCULAR, OPEN OR PERCUTANEOUS,

| 4.2 drug Use of 2 I antihypertensive 4.3 Use of 2 I inihypertensive 4.4 drug Use of 2 I inihypertensive 4.3 Use of 2 I ilipid-lowering drug 4.3 Use of 2 Ilipid-lowering drug 4.3 Use of 2 Ilipid-lowering drug 4.4 Use of 2 I | ICD-10-CM | 4.2 drug Use of 2 I antihypertensive 4.3 drug Use of 2 I antihypertensive 4.4 drug Use of 2 I antihypertensive 4.5 drug Use of 2 I antihypertensive 4.6 drug Use of 2 I antihypertensive 4.7 drug Use of 2 I antihypertensive 4.2 drug Use of 2 I antihypertensive 4.3 Use of 2 I i i i i i i i i i i i i i i i i i i | | Use of ≥ 1 antihypertensive | | | | |
|---|---|---|---|---|---|---|---|---|
| 4.2 drug Use of 2 Intithypertensive 4.3 Use of 2 Intithypertensive 4.3 Use of 2 Ilipid-lowering drug 4.3 Use of 2 Il | Generic | 4.2 drug Use of 1 antihypertensive 4.3 drug Use of 1 antihypertensive 4.4 drug Use of 1 antihypertensive 4.3 drug Use of 1 antihypertensive 4.4 drug Use of 1 antihypertensive 4.3 drug Use of 1 antihypertensive 4.4 drug Use of 1 antihypertensive 4.5 drug Use of 1 antihypertensive 4.6 drug Use of 1 antihypertensive 4.7 drug Use of 1 antihypertensive 4.2 drug Use of 1 antihypertensive 4.3 drug Use of 1 antihypertensive 4.4 drug Use of 1 antihypertensive 4.5 drug Use of 1 antihypertensive 4.6 drug Use of 1 antihypertensive 4.7 drug Use of 1 antihypertensive 4.2 drug Use of 1 antihypertensive 4.3 drug Use of 1 antihypertensive 4.4 drug Use of 1 antihypertensive 4.5 drug Use of 1 antihypertensive 4.6 drug Use of 1 antihypertensive 4.6 drug Use of 1 antihypertensive 4.7 drug Use of 1 antihypertensive 4.2 drug Use of 1 antihypertensive 4.3 Use of 1 lipid-drugening drug 4.3 Use of 1 lipid-dru | 4.2 | drug | LOSARTANPOT | TRX | | Generic |
| 4.2 drug Use of ≥1 antihypertensive 4.3 drug Use of ≥1 inipid-lowering drug 4.3 Use of ≥1 lipid-lowering drug 4.3 | Generic | 4.2 drug Use of ≥1 antihypertensive Use of ≥1 a | | = : | OLMESARTAN | NRX | | Generic |
| Use of ≥ 1 antihypertensive 4.2 drug Use of ≥ 1 antihypertensive 4.3 Use of ≥ 1 antihypertensive 4.3 Use of ≥ 1 lipid-lowering drug 4.4 Use of ≥ 1 lipid-lowering dr | Generic | Use of £ 1 and thypertensive VALSARTAN RX | | | TEL MICA DTAN | DV | | 0 |
| Use of ≥1 antihypertensive 4.2 drug Use of ≥1 antihypertensive 4.3 Use of ≥1 antihypertensive 4.4 drug Use of ≥1 antihypertensive 4.3 Use of ≥1 lipid-lowering drug 4.3 Use of ≥1 lipid-lower | Generic | Use of ≥ 1 antihypertensive All LODIPINE BERX All LODIPINE BERX Generic Use of ≥ 1 antihypertensive LODIPINE BERX LODIP | | 9 | TELMISARTAN | KX | | Generic |
| 4.2 drug Use of ≥1 antihypertensive 4.3 Use of ≥1 lipid-lowering drug 4.3 Use of ≥1 l | Generic | 4.2 drug Use of 2 Intilhypertensive 4.3 Use of 2 Intilhypertensive 4.4 drug Use of 2 Intilhypertensive 4.4 drug Use of 2 Intilhypertensive 4.5 drug 2 Intilhypertensive 4.5 d | | 9 | VALSARTAN | RX | | Generic |
| 4.2 drug Use of ≥1 antihypertensive 4.3 drug Use of ≥1 antihypertensive 4.3 Use of ≥1 lipid-lowering drug 4.3 Use of ≥1 lipid | Generic | 4.2 drog Use of 21 antithypertensive ALL DOTRINE BE RX Generic 4.2 drog Use of 21 antithypertensive KICARDIPINE HURX Generic 4.2 drog Use of 21 antithypertensive MICARDIPINE HURX Generic 4.2 drog Use of 21 antithypertensive MISCOLIPINE RX Generic 4.2 drog Use of 21 antithypertensive Use of 21 antithypertensive Use of 21 antithypertensive Ceneric Ceneric 4.3 Use of 21 lipid-lowering drug Use of 22 lipid-lowering drug Use of 22 lipid-lowering drug Use of 22 lipid-lowering drug Use of 22 lipid-lowering drug Us | 4.2 | drug | AMLODIPINE BE | ERX | | Generic |
| Use of ≥1 antihypertensive 4.2 drug Use of ≥1 antihypertensive 4.3 drug Use of ≥1 antihypertensive 4.3 drug Use of ≥1 antihypertensive 4.3 drug Use of ≥1 antihypertensive 4.3 drug Use of ≥1 antihypertensive 4.3 Use of ≥1 lipid-lowering drug 4.4 Use of ≥1 lipid-lowering drug 4.5 Use of ≥1 lipid-lowering drug 4.6 Use of ≥1 lipid-lowering drug 4.7 Use of ≥1 lipid-lowering drug 4.8 Use of ≥1 lipid-lowering drug 4.9 Use of ≥1 lipid-lowering drug 4.0 Use of ≥1 lipid-lowering drug 4.1 Use of ≥1 lipid-lowering drug 4.2 Use of ≥1 lipid-lowering drug 4.3 Use of ≥1 lipid-lowering drug 4.4 Use of ≥1 lipid-lowering drug 4.5 Use of ≥1 lipid-lowering drug 4.6 Use of ≥1 lipid-lowering drug 4.7 Use of ≥1 lipid- | Generic | Use of \$1 antihypertensive | | | AMLODIPINE BE | ERX | | Generic |
| Use of ≥ 1 antihypertensive 4.2 drug Use of ≥ 1 antihypertensive 4.3 use of ≥ 1 lipid-lowering drug 4.3 Use of ≥ 1 lipid-lowering drug 4.4 Use of ≥ 1 lipid-lowering drug 4.5 Use of ≥ 1 lipid-lowering drug 4.6 Use of ≥ 1 lipid-lowering drug 4.7 Use of ≥ 1 lipid-lowering drug 4.8 Use of ≥ 1 lipid-lowering drug 4.9 Use of ≥ 1 lipid-lowering drug 4.1 Use of ≥ 1 lipid-lowering drug 4.2 Use of ≥ 1 lipid-lowering drug 4.3 Use of ≥ 1 lipid-lowering drug 4.4 Use of ≥ 1 lipid-lowering drug 4.5 Use of ≥ 1 lipid-lowering drug 4.6 Use of ≥ 1 lipid-lowering drug 4.7 Use of ≥ 1 lipid-lowering drug 4.8 Use of ≥ 1 lipid-lowering drug 4.9 Use of ≥ 1 lipid-lowering drug 4.0 Use of ≥ 1 lipid-lowering drug 4.1 Use of ≥ 1 lipid-lowering drug 4.2 Use of ≥ 1 lipid-lowering drug 4.3 Use of ≥ 1 lipid-lowering drug 4.4 Use | Generic | Use of 1 antihyportensive 4.2 drug Use of 2 lantihyportensive 4.3 drug of 2 lantihyportensive 4.4 drug Use of 2 lantihyportensive 4.3 drug of 2 lantihyportensive 4.3 dr | | | EEL ODIDINE | DV | | Camania |
| Use of ≥ 1 antihypertensive 4.2 drug Use of ≥ 1 antihypertensive 4.2 drug Use of ≥ 1 antihypertensive 4.2 drug Use of ≥ 1 antihypertensive 4.2 drug Use of ≥ 1 antihypertensive 4.2 drug Use of ≥ 1 antihypertensive 4.3 drug Use of ≥ 1 antihypertensive 4.4 drug Use of ≥ 1 antihypertensive 4.5 drug Use of ≥ 1 antihypertensive 4.6 drug Use of ≥ 1 antihypertensive 4.7 drug Use of ≥ 1 antihypertensive 4.8 drug Use of ≥ 1 antihypertensive 4.9 drug Use of ≥ 1 antihypertensive 4.1 drug Use of ≥ 1 antihypertensive 4.2 drug Use of ≥ 1 antihypertensive 4.3 Use of ≥ 1 antihypertensive 4.4 drug Use of ≥ 1 antihypertensive 4.5 drug Use of ≥ 1 antihypertensive 4.6 drug Use of ≥ 1 antihypertensive 4.7 drug Use of ≥ 1 antihypertensive 4.8 drug Use of ≥ 1 antihypertensive 4.9 drug Use of ≥ 1 antihypertensive 4.1 disease History of coronary artery History of coronary artery 4.1 disease History of coronary artery History of coronary artery 4.1 disease History of coronary artery 4.1 disease History of coronary artery History of coronary artery 4.1 disease History of coronary artery History of coronary artery History of coronary artery A.1 disease History of coronary artery History of coronary artery A.1 disease History of coronary artery History of coronary artery A.1 disease History of coronary artery A.2 drug A.3 dr | Generic | Use of 2 antihypertensive 4.2 drug Use of 2 lipid-lowering drug 4.3 Use of 2 lipid-lowering drug PRAYASTATIN SODIUM Generic | | 9 | FELODIPINE | KX | | Generic |
| Use of ≥1 antihypertensive 4.2 drug Use of ≥1 antihypertensive 4.2 drug Use of ≥1 antihypertensive 4.2 drug Use of ≥1 antihypertensive 4.2 drug Use of ≥1 antihypertensive 4.2 drug Use of ≥1 antihypertensive 4.3 drug Use of ≥1 antihypertensive 4.4 drug Use of ≥1 antihypertensive 4.3 Use of ≥1 lilpid-lowering drug 4.4 Use of ≥1 lilpid-lowering drug 4.5 Use of ≥1 lilpid-lowering drug 4.6 Use of ≥1 lilpid-lowering drug 4.7 Use of ≥1 lilpid-lowering drug 4.8 Use of ≥1 lilpid-lowering drug 4.9 Use of ≥1 lilpid-lowering drug 4.0 Use of ≥1 lilpid-lowering drug 4.1 disease 4.2 Use of ≥1 lilpid-lowering drug 4.3 Use of ≥1 lilpid-lowering drug 4.4 Use of ≥1 lilpid-lowering drug 4.5 Use of ≥1 lilpid-lowering drug 4.6 Use of ≥1 lilpid-lowering drug 4.7 Use of ≥1 lilpid-lowering drug 4.8 Use of ≥1 lilpid-lowering drug 4.9 Use of ≥1 lilpid-lowering drug 4.0 Use of ≥1 lilpid-lowering drug 4.1 disease 4.2 Use of ≥1 lilpid-lowering drug 4.3 Use of ≥1 lilpid-lowering drug 4.4 Use of ≥1 lilpid-lowering drug 4.5 Use of ≥1 lilpid-lowering drug 4.6 Use of ≥1 lilpid-loweri | Generic | 4.2 drug Use of ≥1 antihypertensive 4.2 drug Use of ≥1 antihypertensive 4.2 drug Use of ≥1 antihypertensive 4.2 drug Use of ≥1 antihypertensive 4.2 drug Use of ≥1 antihypertensive 4.3 drug Use of ≥1 antihypertensive 4.3 drug Use of ≥1 antihypertensive 4.3 use of ≥1 lipid-lowering drug 4.3 Use of ≥1 lipid-lower | | | NICARDIPINE H | (RX | | Generic |
| 4.2 drug Use of ≥1 antihypertensive 4.2 drug Use of ≥1 antihypertensive 4.2 drug Use of ≥1 antihypertensive 4.2 drug Use of ≥1 lipid-lowering drug 4.3 Use of ≥1 lipid-lowering | Generic | A2 drug | 4.2 | drug | NIFEDIPINE | RX | | Generic |
| 4.2 drug Useof≥1 antihypertensive 4.2 drug Useof≥1 antihypertensive 4.2 drug Useof≥1 lipid-lowering drug VERAPAMIL HC RX ATORVASTATIN CALCIUM FLUVASTATIN SODIUM LOVASTATIN LOVAS | Generic | 4.2 drug Use of ≥1 antihypertensive 4.2 drug Use of ≥1 antihypertensive 4.2 drug Use of ≥1 antihypertensive 4.2 drug VERAPAMIL HC RX Generic | | | NISOLDIPINE | RX | | Generic |
| Use of ≥ 1 antihypertensive 4.2 drug 4.3 Use of ≥ 1 lipid-lowering drug 4.4 Use of ≥ 1 lipid-lowering drug 4.5 Use of ≥ 1 lipid-lowering drug 4.6 Use of ≥ 1 lipid-lowering drug 4.7 Use of ≥ 1 lipid-lowering drug 4.8 Use of ≥ 1 lipid-lowering drug 4.9 Use of ≥ 1 lipid-lowering drug 4.1 Use of ≥ 1 lipid-lowering drug 4.2 Use of ≥ 1 lipid-lowering drug 4.3 Use of ≥ 1 lipid-lowering drug 4.4 Use of ≥ 1 lipid-lowering drug 4.5 Use of ≥ 1 lipid-lowering drug 4.6 Use of ≥ 1 lipid-lowering drug 4.7 Use of ≥ 1 lipid-lowering drug 4.8 Use of ≥ 1 lipid-lowering drug 4.9 Use of ≥ 1 lipid-lowering drug 4.1 Use of ≥ 1 lipid-lowering drug 4.2 Use of ≥ 1 lipid-lowering drug 4.3 Use of ≥ 1 lipid-lowering drug 4.4 Use of ≥ 1 lipid-lowering drug 4.5 Use of ≥ 1 lipid-lowering drug 4.6 Use of ≥ 1 lipid-lowering drug 4.7 Use of ≥ 1 lipid-lowering drug 4.8 Use of ≥ 1 lipid-lowering drug 4.9 Use of ≥ 1 lipid-lowering drug 4.1 Use of ≥ 1 lipid-lowering drug 4.2 Use of ≥ 1 lipid-lowering drug 4.3 Use of ≥ 1 lipid-lowering drug 4.4 Use of ≥ 1 lipid-lowering drug 4.5 Use of ≥ 1 lipid-lowering drug 4.6 Use of ≥ 1 lipid-lowering drug 4.7 Use of ≥ 1 lipid-lowering drug 4.8 Use of ≥ 1 lipid-lowering drug 4.9 Use of ≥ | Generic | Use of ≥ 1 antihypertensive 1.2 drug Use of ≥ 1 antihypertensive 1.2 drug Use of ≥ 1 antihypertensive 1.3 Use of ≥ 1 lipid-lowering drug 1.3 Use of ≥ 1 | | = : | | | | |
| 4.2 drug Use of ≥1 antihypertensive 4.2 drug 4.3 Use of ≥1 lipid-lowering drug 4.4 Use of ≥1 lipid-lowering drug 4.5 Use of ≥1 lipid-lowering drug 4.6 Use of ≥1 lipid-lowering drug 4.7 Use of ≥1 lipid-lowering drug 4.8 Use of ≥1 lipid-lowering drug 4.9 Use of ≥1 lipid-lowering drug 4.1 Use of ≥1 lipid-lowering drug 4.2 Use of ≥1 lipid-lowering drug 4.3 Use of ≥1 lipid-lowering drug 4.4 Use of ≥1 lipid-lowering drug 4.5 Use of ≥1 lipid-lowering drug 4.6 Use of ≥1 lipid-lowering drug 4.7 Use of ≥1 lipid-lowering drug 4.8 Use of ≥1 lipid-lowering drug 4.9 Use of ≥1 lipid-lowering drug 4.1 Use of ≥1 lipid-lowering drug 4.2 Use of ≥1 lipid-lowering drug 4.3 Use of ≥1 lipid-lowering drug 4.4 Use of ≥1 lipid-lowering drug 4.5 Use of ≥1 lipid-lowering drug 4.6 Use of ≥1 lipid-lowering drug 4.7 Use of ≥1 lipid-lowering drug 4.8 Use of ≥1 lipid-lowering drug 4.9 Use of ≥1 lipid-lowering drug 4.1 Use of ≥1 lipid-lowering drug 4.2 Use of ≥1 lipid-lowering drug 4.3 Use of ≥1 lipid-lowering drug 4.4 Use of ≥1 lipid-lowering drug 4.5 Use of ≥1 lipid-lowering drug 4.6 Use of ≥1 lipid-lowering drug 4.7 Use of ≥1 lipid-lowering drug 4.8 Use of ≥1 lipid-lowering drug 4.9 Use of ≥1 lipid-lowering drug 4.1 Use of ≥1 lipid-lowering drug 4.2 Use of ≥1 lipid-lowering drug 4.3 Use of ≥1 lipid-lowerin | Generic | 4.2 drug Use of ≥ 1 antihypertensive 4.2 drug 4.3 Use of ≥ 1 lipid-lowering | | 9 | DILTIAZEM HCL | _RX | | Generic |
| 4.2 drug 4.3 Useof≥1lipid-lowering drug 4.4 Useof≥1lipid-lowering drug 4.5 Useof≥1lipid-lowering drug 4.6 Useof≥0 | Generic | 4.2 drug 4.3 Useof≥1lipid-lowering drug 4.4 Useose 4.5 Useof≥1lipid-lowering drug 4.6 Useose 4.7 Useose 4.8 Useose 4.9 Useose 4.1 Useose 4.1 Useose 4.1 Useose 4.2 Useose 4.3 Useof≥1lipid-lowering drug 4.4 Useose 4.4 Useose 4.5 Useose 4.6 Useose 4.6 Useose 4.7 Useose 4.8 Useose 4.8 Useose 4.9 Useose 4.9 Useose 4.1 Useose 4.1 Useose 4.1 Useose 4.2 Useose 4.3 Useose 4.4 Useose | 4.2 | drug | DILTIAZEM MAL | LRX | | Generic |
| 4.3 Use of≥1 lipid-lowering drug 4.4 Use accordance drug 4.5 Use of≥1 lipid-lowering drug 4.6 Use accordance drug 4.7 Use accordance drug 4.8 Use of≥1 lipid-lowering drug 4.9 Use of≥1 lipid-lowering drug 4.1 Use accordance drug 4.2 Use of≥1 lipid-lowering drug 4.3 Use of≥1 lipid-lowering drug 4.4 Use accordance drug 4.5 Use of≥1 lipid-lowering drug 4.6 Use accordance drug 4.7 Use accordance drug 4.8 Use of≥1 lipid-lowering drug 4.9 Use of≥1 lipid-lowering drug 4.1 Use accordance drug 4.2 Use of≥1 lipid-lowering drug 4.3 Use of≥1 lipid-lowering drug 4.4 Use accordance drug 4.5 Use of≥1 lipid-lowering drug 4.6 Use accordance drug 4.7 Use accordance drug 4.8 Use of≥1 lipid-lowering drug 4.9 Use of≥1 lipid-lowering drug 4.1 Use accordance drug 4.2 Use of≥1 lipid-lowering drug 4.3 Use of≥1 lipid-lowering drug 4.4 Use accordance drug 4.5 Use of≥1 lipid-lowering drug 4.6 Use accordance drug 4.7 Use accordance drug 4.8 Use of≥1 lipid-lowering drug 4.9 Use of≥1 lipid-lowering drug 4.1 Use of≥1 lipid-lowering drug 4.2 Use of≥1 lipid-lowering drug 4.3 Use of≥1 lipid-lowering drug 4.4 Use of≥1 lipid-lowering drug 4.5 Use of≥1 lipid-lowering drug 4.6 Use of≥1 lipid-lowering drug 4.7 Use of≥1 lipid-lowering drug 4.8 Use of≥1 lipid-lowering drug 4.9 Use of≥1 lipid-lowering drug 4.1 Use of≥1 lipid-lowering drug 4. | Generic | 4.3 Use of 2 Ilipid-lowering drug 4.4 Use ase 4.3 Use of 2 Ilipid-lowering drug 4.4 Use ase 4.4 Use ase 4.5 Use of 2 Ilipid-lowering drug 4.6 Use ase 4.7 Use ase 4.8 Use of 2 Ilipid-lowering drug 4.9 Use of 2 Ilipid-lowering drug 4.1 disease 4.2 Use of 2 Ilipid-lowering drug 4.3 Use of 2 Ilipid-lowering drug 4.4 Use ase 4.5 Use of 2 Ilipid-lowering drug 4.6 Use ase 4.7 Use ase 4.8 Use of 2 Ilipid-lowering drug 4.9 Use of 2 Ilipid-lowering drug 4.1 disease 4.2 Use of 2 Ilipid-lowering drug 4.3 Use of 2 Ilipid-lowering drug 4.4 Use ase 4.5 Use of 2 Ilipid-lowering drug 4.6 Use ase 4.7 Use of 2 Ilipid-lowering drug 4.8 Use of 2 Ilipid-lowering drug 4.9 Use of 2 Ilipid-lowering drug 4.1 disease 4.2 Use of 2 Ilipid-lowering drug 4.3 Use of 2 Ilipid-lowering drug 4.4 Use ase 4.5 Use of 2 Ilipid-lowering drug 4.6 Use of 2 Ilipid-lowering drug 4.7 Use | | 3. | VEDADAMII HO | ` DV | | Conorio |
| 4.3 Use of≥1 lipid-lowering drug 4.4 Use of≥1 lipid-lowering drug 4.5 Use of≥1 lipid-lowering drug 4.6 Use of≥1 lipid-lowering drug 4.7 Use of≥1 lipid-lowering drug 4.8 Use of≥1 lipid-lowering drug 4.9 Use of≥1 lipid-lowering drug 4.1 disease 4.1 disease 4.2 Use of≥1 lipid-lowering drug 4.3 Use of≥1 lipid-lowering drug 4.4 Use of≥1 lipid-lowering drug 4.5 Use of≥1 lipid-lowering drug 4.6 Use of≥1 lipid-lowering drug 4.7 Use of≥1 lipid-lowering drug 4.8 Use of≥1 lipid-lowering drug 4.9 Use of≥1 lipid-lowering drug 4.1 disease 4.2 Use of≥1 lipid-lowering drug 4.3 Use of≥1 lipid-lowering drug 4.4 Use of≥1 lipid-lowering drug 4.5 Use of≥1 lipid-lowering drug 4.6 Use of≥1 lipid-lowering drug 4.7 Use of≥1 lipid-lowering drug 4.8 Use of≥1 lipid-lowering drug 4.9 Use of≥1 lipid-lowering drug 4.1 disease 4.2 Use of≥1 lipid-lowering drug 4.3 Use of≥1 lipid-lowering drug 4.4 Use of≥1 lipid-lowering drug 4.5 Use of≥1 lipid-lowering drug 4.6 Use of≥1 lipid-lowering drug 4.7 Use of≥1 lipid-lowering drug 4.8 Use of≥1 lipid-lowering drug 4.9 Use of≥1 lipid-lowering drug 4.1 disease 4.2 Use of≥1 lipid-lowering drug 4.3 Use of≥1 lipid-lowering drug 4.4 Use of≥1 lipid-lowering drug 4.5 Use of≥1 lipid-lowering drug 4.6 Use of≥1 lipid-lowering drug 4.7 Use of≥1 lipid-lowering drug 4.8 Use of≥1 lipid-lowering drug 4.9 Use of≥1 lipid-lowering drug 4.1 Use of≥1 lipid-lowering drug 4.2 Use of≥1 lipid-lowering drug 4.3 U | Generic | 4.3 Use of 21 lipid-lowering drug 4.4 Use of 21 lipid-lowering drug 4.5 Use of 21 lipid-lowering drug 4.6 Use of 21 lipid-lowering drug 4.7 Use of 21 lipid-lowering drug 4.8 Use of 21 lipid-lowering drug 4.9 Use of 21 lipid-lowering drug 4.1 Use of 21 lipid-lowering drug 4.2 Use of 21 lipid-lowering drug 4.3 Use of 21 lipid-lowering drug 4.4 Use of 21 lipid-lowering drug 4.5 Use of 21 lipid-lowering drug 4.6 Use of 21 lipid-lowering drug 4.7 Use of 21 lipid-lowering drug 4.8 Use of 21 lipid-lowering drug 4.9 Use of 21 lipid-lowering drug 4.1 Use of 21 lipid-lowering drug 4.2 Use of 21 lipid-lowering drug 4.3 Use of 21 lipid-lowering drug 4.4 Use of 21 lipid-lowering drug 4.5 Use of 21 lipid-lowering drug 4.6 Use of 21 lipid-lowering drug 4.7 Use of 21 lipid-lowering drug 4.8 Use of 21 lipid-lowering drug 4.9 Use of 21 lipid-lowering drug 4.1 Use of 21 lipid-lowering drug 4.2 Use of 21 lipid-lowering drug 4.3 Use of 21 lipid-lowering drug 4.4 Use of 21 lipid-lowering drug 4.5 Use of 21 lipid-lowering drug 4.6 Use of 21 lipid-lowering drug 4.7 Use of 21 lipid-lowering drug 4.8 Use of 21 lipid-lowering drug 4.9 Use of 21 lipid-lowering drug 4.1 Use of 21 lipid-lowering drug 4.2 Use of 21 lipid-lowering drug 4.3 Use of 21 lipid-lowering drug 4.4 Use of 21 lipid-lowering drug 4.5 Us | | | | | | |
| 4.3 Use of ≥1 lipid-lowering drug 4.4 Use of ≥1 lipid-lowering drug 4.5 Use of ≥1 lipid-lowering drug 4.6 Use of ≥1 lipid-lowering drug 4.7 Use of ≥1 lipid-lowering drug 4.8 Use of ≥1 lipid-lowering drug 4.9 Use of ≥1 lipid-lowering drug 4.1 disease 4.2 Use of ≥1 lipid-lowering drug 4.3 Use of ≥1 lipid-lowering drug 4.4 Use of ≥1 lipid-lowering drug 4.5 Use of ≥1 lipid-lowering drug 4.6 Use of ≥1 lipid-lowering drug 4.7 Use of ≥1 lipid-lowering drug 4.8 Use of ≥1 lipid-lowering drug 4.9 Use of ≥1 lipid-lowering drug 4.1 Use of ≥1 lipid-lowering drug 4.3 Use of ≥1 lipid-lowering drug 4.4 Use of ≥1 lipid-lowering drug 4.5 Use of ≥1 lipid-lowering drug 4.6 Use of ≥1 lipid-lowering drug 4.7 Use of ≥1 lipid-lowering drug 4.8 Use of ≥1 lipid-lowering drug 4.9 Use of ≥1 lipid-lowering drug 4.1 Use of ≥1 lipid-lowering drug 4.2 Use of ≥1 lipid-lowering drug 4.3 Use of ≥1 lipid-lowering drug 4.4 Use of ≥1 lipid-lowering drug 4.5 Use of ≥1 lipid-lowering drug 4.6 Use of ≥1 lipid-lowering drug 4.8 Use of ≥1 lipid-lowering drug 4.9 Use of ≥1 lipid-lowering drug 4.1 Use of ≥1 lipid-lowering drug 4.2 Use of ≥1 lipid-lowering drug 4.3 Use of ≥1 lipid-lowerin | Generic | 4.3 Use of ≥1 lipid-lowering drug 4.4 Use of ≥1 lipid-lowering drug 4.5 Use of ≥1 lipid-lowering drug 4.6 Use of ≥1 lipid-lowering drug 4.7 Use of ≥1 lipid-lowering drug 4.8 Use of ≥1 lipid-lowering drug 4.9 Use of ≥1 lipid-lowering drug 4.1 Use of ≥1 lipid-lowering drug 4.2 Use of ≥1 lipid-lowering drug 4.3 Use of ≥1 lipid-lowering drug 4.4 Use of ≥1 lipid-lowering drug 4.5 Use of ≥1 lipid-lowering drug 4.6 Use of ≥1 lipid-lowering drug 4.7 Use of ≥1 lipid-lowering drug 4.8 Use of ≥1 lipid-lowering drug 4.9 Use of ≥1 lipid-lowering drug 4.1 Use of ≥1 lipid-lowering drug 4.2 Use of ≥1 lipid-lowering drug 4.3 Use of ≥1 lipid-lowering drug 4.4 Use of ≥1 lipid-lowering drug 4.4 Use of ≥1 lipid-lowering drug 4.4 Use of ≥1 lipid-lowering drug 4.4 Use of ≥1 lipid-lowering drug 4.5 Use of ≥1 lipid-lowering drug 4.6 Use of ≥1 lipid-lowering drug 4.7 Use of ≥1 lipid-lowering drug 4.8 Use of ≥1 lipid-lowering drug 4.9 Use of ≥1 lipid-lowering drug 4.1 Use of ≥1 lipid-lowering drug 4.2 Use of ≥1 lipid-lowering drug 4.3 Use of ≥1 lipid-lowering drug 4.4 Use of ≥1 lipid-lowering drug 4.5 Use of ≥1 lipid-lowering drug 4.6 Use of ≥1 lipid-lowering drug 4.7 Use of ≥1 lipid-lowering drug 4.8 Use of ≥1 lipid-lowering drug 4.9 Use of ≥1 lipid-lowering drug 4.1 Use of ≥1 lipid-lowering drug 4.2 Use of ≥1 lipid-lowering drug 4.3 Use of ≥1 lipid-lowering drug 4.4 Use of ≥1 lipid-lowering drug 4.5 U | | | | | | |
| 4.3 Use of ≥ 1 lipid-lowering drug 4.4 Use of ≥ 1 lipid-lowering drug 4.5 Use of ≥ 1 lipid-lowering drug 4.6 Use of ≥ 1 lipid-lowering drug 4.7 Use of ≥ 1 lipid-lowering drug 4.8 Use of ≥ 1 lipid-lowering drug 4.9 Use of ≥ 1 lipid-lowering drug 4.1 disease 4.2 Use of ≥ 1 lipid-lowering drug 4.3 Use of ≥ 1 lipid-lowering drug 4.4 Use of ≥ 1 lipid-lowering drug 4.5 Use of ≥ 1 lipid-lowering drug 4.6 Use of ≥ 1 lipid-lowering drug 4.7 Use of ≥ 1 lipid-lowering drug 4.8 Use of ≥ 1 lipid-lowering drug 4.9 Use of ≥ 1 lipid-lowering drug 4.1 disease 4.2 Use of ≥ 1 lipid-lowering drug 4.3 Use of ≥ 1 lipid-lowering drug 4.4 Use of ≥ 1 lipid-lowering drug 4.5 Use of ≥ 1 lipid-lowering drug 4.6 Use of ≥ 1 lipid-lowering drug 4.7 Use of ≥ 1 lipid-lowering drug 4.8 Use of ≥ 1 lipid-lowering drug 4.9 Use of ≥ 1 lipid-lowering drug 4.1 disease 4.2 Use of ≥ 1 lipid-lowering drug 4.3 Use of ≥ 1 lipid-lowering drug 4.4 Use of ≥ 1 lipid-lowering drug 4.5 Use of ≥ 1 lipid-lowering drug 4.6 Use of ≥ 1 lipid-lowering drug 4.7 Use of ≥ 1 lipid-lowering drug 4.8 Use of ≥ 1 lipid-lowering drug 4.9 Use of ≥ 1 lipid-lowering drug 4.1 disease 4.2 Use of ≥ 1 lipid-lowering drug 4.3 Use of ≥ 1 lipid-lowering drug 4. | Generic | 4.3 Use of ≥ 1 lipid-lowering drug PITAVASTATIN CALCIUM Generic 4.3 Use of ≥ 1 lipid-lowering drug PITAVASTATIN MAGNESIUM Generic 4.3 Use of ≥ 1 lipid-lowering drug PITAVASTATIN SODIUM Generic 4.3 Use of ≥ 1 lipid-lowering drug ROSUVASTATIN CALCIUM Generic 4.3 Use of ≥ 1 lipid-lowering drug CHOLESTYRAMINE Generic 4.3 Use of ≥ 1 lipid-lowering drug CHOLESTYRAMINE Generic 4.3 Use of ≥ 1 lipid-lowering drug COLESTUPOL HCL Generic 4.3 Use of ≥ 1 lipid-lowering drug EVOLOCUMAB Generic 4.3 Use of ≥ 1 lipid-lowering drug EVOLOCUMAB Generic 4.3 Use of ≥ 1 lipid-lowering drug EVOLOCUMAB Generic 4.3 Use of ≥ 1 lipid-lowering drug EVOLOCUMAB Generic 4.3 Use of ≥ 1 lipid-lowering drug EVOLOCUMAB Generic 4.3 Use of ≥ 1 lipid-lowering drug EVOLOCUMAB Generic 4.3 Use of ≥ 1 lipid-lowering drug EVOLOCUMAB Generic 4.3 Use of ≥ 1 lipid-lowering drug EVOLOCUMAB Generic 4.4.1 disease ISOLOCUMAB ISOLOCUMAB ISOLOCUMAB </th <th></th> <th></th> <th></th> <th>30210111</th> <th></th> <th></th> | | | | 30210111 | | |
| 4.3 Use of≥1 lipid-lowering drug 4.4 Use of≥1 lipid-lowering drug 4.5 Use of≥1 lipid-lowering drug 4.6 Use of≥1 lipid-lowering drug 4.7 Use of≥1 lipid-lowering drug 4.8 Use of≥1 lipid-lowering drug 4.9 Use of≥1 lipid-lowering drug 4.1 disease History of coronary artery | Generic | 4.3 Use of ≥1 lipid-lowering drug 4.4 Use as of ≥1 lipid-lowering drug 4.5 Use of ≥1 lipid-lowering drug 4.6 Use of ≥1 lipid-lowering drug 4.7 Use of ≥1 lipid-lowering drug 4.8 Use of ≥1 lipid-lowering drug 4.9 Use of ≥1 lipid-lowering drug 4.1 Use as of ≥1 lipid-lowering drug 4.2 Use of ≥1 lipid-lowering drug 4.3 Use of ≥1 lipid-lowering drug 4.4 Use as of ≥1 | | | | CALCIUM | | |
| 4.3 Use of≥1 lipid-lowering drug 4.4 Use of≥1 lipid-lowering drug History of coronary artery 4.4.1 disease History of coronary artery | Generic ICD-10-CM ICD-10-CM | 4.3 Use of ≥1 lipid-lowering drug 4.4 Use of ≥1 lipid-lowering drug 4.5 Use of ≥1 lipid-lowering drug 4.6 Use of ≥1 lipid-lowering drug 4.7 Use of ≥1 lipid-lowering drug 4.8 Use of ≥1 lipid-lowering drug 4.9 Use of ≥1 lipid-lowering drug 4.1 disease History of coronary artery 4.1 disease History of coronary artery 4.1 disease History of coronary artery 4.1 disease Uso 9 DX Angina pectoris with coronary microvascular dysfunction Uso 10-10-CM History of coronary artery 4.1 disease Lipid-lowering drug History of coronary artery 4.1 disease History of coronary artery 4.1 disease History of coronary artery 4.1 disease Lipid-lowering drug History of coronary artery 4.1 disease History of coronary artery 4.1 disease Lipid-lowering drug History of coronary artery Angle Period Roberts History of coronary | | | | | | |
| 4.3 Use of≥1lipid-lowering drug 4.4 Use of≥1lipid-lowering drug History of coronary artery 4.4.1 disease History of coronary artery | Generic HCD-10-CM HCD-10-CM HCD-10-CM | 4.3 Use of ≥1 lipid-lowering drug History of coronary artery 4.4.1 disease History of coronary artery 4.4.2 disease History of coronary artery 4.4.3 disease History of coronary artery 4.4.4 disease History of coronary artery 4.4.5 disease History of coronary artery 4.4.6 disease History of coronary artery 4.4.7 disease History of coronary artery 4.4.8 disease History of coronary artery 4.4.9 disease History of coronary artery 4.4.1 disease History of coronary artery 4.4.2 disease History of coronary artery 4.4.3 disease History of coronary artery 4.4.4 disease History of coronary artery 4.5 disease History of coronary artery 4.6 disease H | | | | | | |
| 4.3 Use of ≥1 lipid-lowering drug History of coronary artery 4.4.1 disease History of coronary artery | Generic ICD-10-CM ICD-10-CM ICD-10-CM | 4.3 Use of≥1 lipid-lowering drug History of coronary artery 4.4.1 disease L20.8 DX Angina pectoris with coronary microvascular dysfunction ICD-10-CM History of coronary artery 4.4.1 disease L20.8 DX ANGINA PECTORIS WITH DOCUMENTED SPASM ICD-10-CM History of coronary artery 4.4.1 disease History of coronary artery 4.4.2 disease History of coronary artery 4.4.3 disease History of coronary artery 4.4.4 disease | | | | | | |
| 4.3 Use of ≥1 lipid-lowering drug History of coronary artery 4.4.1 disease I20.0 DX Unstable angina History of coronary artery 4.4.1 disease I20.2 DX Refractory angina pectoris History of coronary artery 4.4.1 disease I20.81 DX Angina pectoris with coronary microvascular dysfunction History of coronary artery 4.4.1 disease I20.89 DX Other forms of angina pectoris History of coronary artery 4.4.1 disease I20.1 DX ANGINA PECTORIS WITH DOCUMENTED SPASM History of coronary artery | Generic ICD-10-CM ICD-10-CM ICD-10-CM | 4.3 Use of ≥1 lipid-lowering drug History of coronary artery 4.1 disease History of coronary artery 4.1 disease I20.0 DX Unstable angina ICD-10-CM History of coronary artery 4.1 disease I20.2 DX Refractory angina pectoris ICD-10-CM History of coronary artery 4.1 disease I20.81 DX Angina pectoris with coronary microvascular dysfunction ICD-10-CM History of coronary artery 4.1 disease I20.89 DX Other forms of angina pectoris History of coronary artery 4.1 disease I20.1 DX ANGINA PECTORIS WITH DOCUMENTED SPASM ICD-10-CM History of coronary artery 4.1 disease I20.8 DX OTHER FORMS OF ANGINA PECTORIS History of coronary artery 4.1 disease I20.9 DX ANGINA PECTORIS, UNSPECIFIED History of coronary artery 4.1 disease I20.9 DX ANGINA PECTORIS WITH DOCUMENTED SPASM ICD-10-CM History of coronary artery 4.1 disease I20.9 DX ANGINA PECTORIS, UNSPECIFIED History of coronary artery 4.1 disease I20.9 DX ANGINA PECTORIS WITH DOCUMENTED SPASM ICD-10-CM History of coronary artery ATHEROSCLEROTIC HEART DISEASE OF NATIVE CORONARY ARTERY History of coronary artery ATHEROSCLEROTIC HEART DISEASE OF NATIVE CORONARY ARTERY | | | | NCALCIUM | | |
| 4.3 Use of ≥1 lipid-lowering drug 4.4 Use of ≥1 lipid-lowering drug 4.5 Use of ≥1 lipid-lowering drug 4.6 Use of ≥1 lipid-lowering drug 4.7 Use of ≥1 lipid-lowering drug 4.8 Use of ≥1 lipid-lowering drug 4.9 Use of ≥1 lipid-lowering drug 4.1 disease 4.2 Use of ≥1 lipid-lowering drug 4.3 Use of ≥1 lipid-lowering drug 4.4 Use of ≥1 lipid-lowering drug 4.5 Use of ≥1 lipid-lowering drug 4.6 Use of ≥1 lipid-lowering drug 4.7 Use of ≥1 lipid-lowering drug 4.8 Use of ≥1 lipid-lowering drug 4.4 Use of ≥1 lipid-lowering drug 4.4 Use of ≥1 lipid-lowering drug 4.4 Use of ≥1 lipid-lowering drug 4.5 Use of ≥1 lipid-lowering drug 4.6 Use of ≥1 lipid-lowering drug 4.7 Use of ≥1 lipid-lowering drug 4.8 Use of ≥1 lipid-lowering drug 4.9 Use of ≥1 lipid-lowering drug 4.4 Use of ≥1 lipid-lowerin | Generic ICD-10-CM ICD-10-CM ICD-10-CM | 4.3 Use of≥1 lipid-lowering drug 4.4 Use of≥1 lipid-lowering drug 4.5 Use of≥1 lipid-lowering drug 4.6 Use of≥1 lipid-lowering drug 4.7 Use of≥1 lipid-lowering drug 4.8 Use of≥1 lipid-lowering drug 4.9 Use of≥1 lipid-lowering drug 4.9 Use of≥1 lipid-lowering drug 4.1 Use of≥1 lipid-lowering drug 4.2 Use of≥1 lipid-lowering drug 4.3 Use of≥1 lipid-lowering drug 4.4 Use of≥1 lipid-lowering drug 5 of or onary artery 4.4 Use of≥1 lipid-lowering drug 6 of onaric 6 of | | | | | | |
| 4.3 Use of ≥1 lipid-lowering drug 4.4 Use of ≥1 lipid-lowering drug History of coronary artery 4.4.1 disease History of coronary artery | Generic Generic Generic Generic Generic ICD-10-CM ICD-10-CM ICD-10-CM ICD-10-CM | 4.3 Use of ≥1 lipid-lowering drug 4.3 Use of ≥1 lipid-lowering drug 4.3 Use of ≥1 lipid-lowering drug 4.3 Use of ≥1 lipid-lowering drug History of coronary artery 4.4.1 disease History of coronary artery 4.4.1 disease History of coronary artery 4.4.2 disease History of coronary artery 4.4.3 disease History of coronary artery 4.4.4 disease History of coronary artery 4.4.5 disease History of coronary artery 4.4.6 disease History of coronary artery 4.4.1 disease History of coronary artery 4.4.2 disease History of coronary artery 4.4.3 disease History of coronary artery 4.4.4 disease History of coronary artery 4.4.5 disease History of coronary artery 4.4.6 disease History of coronary artery 4.4.7 disease History of coronary artery 4.4.8 disease History of coronary artery 4.4.9 disease History of coronary artery 4.4.1 disease History of coronary artery 4.4.2 disease History of coronary artery 4.4.3 disease History of coronary artery 4.4.4 disease History of coronary artery 4.4.5 disease History of coronary artery 4.4.6 disease History of coronary artery 4.4.7 disease History of coronary artery 4.4.8 disease History of coronary artery 4.4.9 disease History of coronary artery 4.4.1 disease History of coronary artery 4.4.2 disease History of coronary artery 4.4.3 disease History of coronary artery 4.4.4 disease History of coronary artery 4.4.5 disease History of coronary artery 4.4.6 disease History of coronary artery 4.4.7 disease History of coronary artery 4.4.8 disease History of coronary artery 4.4.9 disease History of coronary artery 4.4.1 disease History of coronary artery 4.4.2 disease History of coronary artery 4.4.3 disease History of coronary artery 4.4.4 disease History of coronary artery 4.4.5 disease History of coronary artery 4.4.6 disease History of coronary artery 4.4.7 disease History of coronary artery 4.4.8 disease History of coronary artery 4.4.9 disease History of coronary artery 4.4.1 disease History of coronary artery 4.4.2 disease History of coronary artery 4.4.3 disease History of coronary art | 4.3 | Use of ≥1 lipid-lowering drug | CHOLESTYRAM | IINE | | Generic |
| 4.3 Use of ≥1 lipid-lowering drug 4.3 Use of ≥1 lipid-lowering drug 4.3 Use of ≥1 lipid-lowering drug History of coronary artery 4.4.1 disease History of coronary artery | Generic Generic Generic ICD-10-CM ICD-10-CM ICD-10-CM ICD-10-CM | 4.3 Use of ≥ Ilipid-lowering drug 4.3 Use of ≥ Ilipid-lowering drug History of coronary artery 4.4.1 disease History of coronary artery 4.4.2 disease History of coronary artery 4.4.3 disease History of coronary artery 4.4.4 disease History of coronary artery 4.4.5 disease History of coronary artery 4.4.6 disease History of coronary artery 4.4.7 disease History of coronary artery 4.4.8 disease History of coronary artery 4.4.9 disease History of coronary artery 4.4.1 disease History of coronary artery 4.4.2 disease History of coronary artery 4.4.3 disease History of coronary artery 4.4.4 disease History of coronary artery 4.4.5 disease History of coronary artery 4.4.6 disease History of coronary artery 4.4.7 disease History of coronary artery 4.4.8 disease History of coronary artery 4.4.9 disease History of coronary artery 4.4.1 disease History of coronary artery 4.4.2 disease History of coronary artery 4.4.3 disease History of coronary artery 4.4.4 disease History of coronary artery 4.4.5 disease History of coronary artery 4.4.6 disease History of coronary artery 4.4.7 disease History of coronary artery 4.4.8 disease History of coronary artery 4.4.9 disease History of coronary artery 4.4.1 disease History of coronary artery 4.4.2 disease History of coronary artery 4.4.3 disease History of coronary artery History of coronary artery History of coronary artery History of | 4.3 | Use of ≥1 lipid-lowering drug | COLESEVELAM | IHCL | | Generic |
| 4.3 Use of ≥1 lipid-lowering drug History of coronary artery 4.4.1 disease History of coronary artery | Generic Generic ICD-10-CM ICD-10-CM ICD-10-CM ICD-10-CM | 4.3 Use of≥1lipid-lowering drug History of coronary artery 4.4.1 disease History of coronary artery 4.4.2 disease History of coronary artery 4.4.3 disease History of coronary artery 4.4.4 disease History of coronary artery 4.4.5 disease History of coronary artery 4.4.6 disease History of coronary artery 4.4.7 disease History of coronary artery 4.4.8 disease History of coronary artery 4.4.9 disease History of coronary artery 4.4.1 disease History of coronary artery 4.4.2 disease History of coronary artery 4.4.3 disease History of coronary artery 4.4.4 disease Hist | 4.3 | Use of ≥1 lipid-lowering drug | COLESTIPOL HO | CL | | Generic |
| 4.3 Use of ≥1 lipid-lowering drug History of coronary artery 4.4.1 disease I20.0 DX Unstable angina History of coronary artery 4.4.1 disease I20.2 DX Refractory angina pectoris History of coronary artery 4.4.1 disease I20.81 DX Angina pectoris with coronary microvascular dysfunction History of coronary artery 4.4.1 disease I20.89 DX Other forms of angina pectoris History of coronary artery 4.4.1 disease I20.89 DX ANGINA PECTORIS WITH DOCUMENTED SPASM History of coronary artery | Generic ICD-10-CM ICD-10-CM dysfunction ICD-10-CM ICD-10-CM | 4.3 Use of ≥1 lipid-lowering drug History of coronary arteryEVOLOCUMAB History of coronary arteryGeneric Generic Generic Generic Generic History of coronary artery4.4.1 disease History of coronary arteryIZO.2DXRefractory angina pectorisICD-10-CM Generic | 4.3 | Use of ≥1 lipid-lowering drug | EZETIMIBE | | | Generic |
| History of coronary artery 4.4.1 disease | ICD-10-CM ICD-10-CM dysfunction ICD-10-CM ICD-10-CM | History of coronary artery 4.4.1 disease 120.0 DX Unstable angina ICD-10-CM History of coronary artery 4.4.1 disease 120.2 DX Refractory angina pectoris ICD-10-CM History of coronary artery 4.4.1 disease 120.81 DX Angina pectoris with coronary microvascular dysfunction ICD-10-CM History of coronary artery 4.4.1 disease 120.89 DX Other forms of angina pectoris ICD-10-CM History of coronary artery 4.4.1 disease 120.1 DX ANGINA PECTORIS WITH DOCUMENTED SPASM ICD-10-CM History of coronary artery 4.4.1 disease 120.8 DX OTHER FORMS OF ANGINA PECTORIS ICD-10-CM History of coronary artery 4.4.1 disease 120.9 DX ANGINA PECTORIS, UNSPECIFIED ICD-10-CM History of coronary artery 4.4.1 disease 120.9 DX ANGINA PECTORIS, UNSPECIFIED ICD-10-CM ATHEROSCLEROTIC HEART DISEASE OF NATIVE CORONARY ARTERY 4.4.1 disease 125.111 DX WITH ANGINA PECTORIS WITH DOCUMENTED SPASM ICD-10-CM ATHEROSCLEROTIC HEART DISEASE OF NATIVE CORONARY ARTERY ICD-10-CM | 4.3 | Use of ≥1 lipid-lowering drug | ALIROCUMAB | | | Generic |
| 4.4.1 disease History of coronary artery 4.4.1 disease History of coronary artery 4.4.1 disease History of coronary artery 4.4.1 disease I20.81 DX Angina pectoris with coronary microvascular dysfunction History of coronary artery 4.4.1 disease I20.89 DX Other forms of angina pectoris History of coronary artery 4.4.1 disease I20.1 DX ANGINA PECTORIS WITH DOCUMENTED SPASM History of coronary artery | dysfunction ICD-10-CM ICD-10-CM | 4.4.1 disease I20.0 DX Unstable angina ICD-10-CM History of coronary artery 4.4.1 disease I20.2 DX Refractory angina pectoris ICD-10-CM History of coronary artery 4.4.1 disease I20.81 DX Angina pectoris with coronary microvascular dysfunction ICD-10-CM History of coronary artery 4.4.1 disease I20.89 DX Other forms of angina pectoris ICD-10-CM History of coronary artery 4.4.1 disease I20.1 DX ANGINA PECTORIS WITH DOCUMENTED SPASM ICD-10-CM History of coronary artery 4.4.1 disease I20.8 DX OTHER FORMS OF ANGINA PECTORIS ICD-10-CM History of coronary artery 4.4.1 disease I20.9 DX ANGINA PECTORIS, UNSPECIFIED ICD-10-CM History of coronary artery 4.4.1 disease I20.9 DX ANGINA PECTORIS, UNSPECIFIED ICD-10-CM History of coronary artery 4.4.1 disease I20.9 DX ATHEROSCLEROTIC HEART DISEASE OF NATIVE CORONARY ARTERY 4.4.1 disease I20.9 ICD-10-CM ATHEROSCLEROTIC HEART DISEASE OF NATIVE CORONARY ARTERY 4.4.1 disease I20.9 ICD-10-CM ATHEROSCLEROTIC HEART DISEASE OF NATIVE CORONARY ARTERY 4.4.1 disease I20.9 ICD-10-CM ATHEROSCLEROTIC HEART DISEASE OF NATIVE CORONARY ARTERY 4.4.1 disease I20.9 ICD-10-CM ATHEROSCLEROTIC HEART DISEASE OF NATIVE CORONARY ARTERY | 4.3 | Use of ≥1 lipid-lowering drug | <b>EVOLOCUMAB</b> | | | Generic |
| History of coronary artery 4.4.1 disease I20.2 DX Refractory angina pectoris 4.4.1 disease I20.81 DX Angina pectoris with coronary microvascular dysfunction History of coronary artery 4.4.1 disease I20.89 DX Other forms of angina pectoris History of coronary artery 4.4.1 disease I20.1 DX ANGINA PECTORIS WITH DOCUMENTED SPASM History of coronary artery | dysfunction ICD-10-CM ICD-10-CM | History of coronary artery 4.4.1 disease I20.2 DX Refractory angina pectoris ICD-10-CM History of coronary artery 4.4.1 disease I20.81 DX Angina pectoris with coronary microvascular dysfunction ICD-10-CM History of coronary artery 4.4.1 disease I20.89 DX Other forms of angina pectoris ICD-10-CM History of coronary artery 4.4.1 disease I20.1 DX ANGINA PECTORIS WITH DOCUMENTED SPASM ICD-10-CM History of coronary artery 4.4.1 disease I20.8 DX OTHER FORMS OF ANGINA PECTORIS ICD-10-CM History of coronary artery 4.4.1 disease I20.9 DX ANGINA PECTORIS, UNSPECIFIED ICD-10-CM History of coronary artery 4.4.1 disease I20.9 DX ANGINA PECTORIS, UNSPECIFIED ICD-10-CM ATHEROSCLEROTIC HEART DISEASE OF NATIVE CORONARY ARTERY 4.4.1 disease I25.111 DX WITH ANGINA PECTORIS WITH DOCUMENTED SPASM ICD-10-CM ATHEROSCLEROTIC HEART DISEASE OF NATIVE CORONARY ARTERY ATHEROSCLEROTIC HEART DISEASE OF NATIVE CORONARY ARTERY | | History of coronary artery | | | | |
| 4.4.1 disease History of coronary artery 4.4.1 disease I20.81 DX Angina pectoris with coronary microvascular dysfunction History of coronary artery 4.4.1 disease I20.89 DX Other forms of angina pectoris History of coronary artery 4.4.1 disease I20.1 DX ANGINA PECTORIS WITH DOCUMENTED SPASM History of coronary artery | dysfunction ICD-10-CM ICD-10-CM | 4.4.1 disease History of coronary artery IZO.2 DX Refractory angina pectoris ICD-10-CM Performs of angina pectoris with coronary microvascular dysfunction ICD-10-CM Performs of angina pectoris 4.4.1 disease History of coronary artery IZO.89 DX Other forms of angina pectoris ICD-10-CM Performs of angina pectoris 4.4.1 disease History of coronary artery IZO.1 DX ANGINA PECTORIS WITH DOCUMENTED SPASM ICD-10-CM Performs of ANGINA PECTORIS 4.4.1 disease History of coronary artery IZO.9 DX ANGINA PECTORIS, UNSPECIFIED PECTORIS, UNSPECTORIS, UNSPECIFIED PECTORIS, UNSPECTORIS, UNSPECTORIS, UNSPECTORIS, UNSPECTORIS, UNSPECTORIS, UNSPECTORIS, UNSPECTORIS, UNSPECT | 4.4.1 | disease | 120.0 | DX | Unstable angina | ICD-10-CM |
| History of coronary artery 4.4.1 disease History of coronary artery 4.4.1 disease I20.81 DX Angina pectoris with coronary microvascular dysfunction History of coronary artery 4.4.1 disease I20.89 DX Other forms of angina pectoris History of coronary artery 4.4.1 disease I20.1 DX ANGINA PECTORIS WITH DOCUMENTED SPASM History of coronary artery | dysfunction ICD-10-CM ICD-10-CM | History of coronary artery 4.4.1 disease I20.81 DX Angina pectoris with coronary microvascular dysfunction ICD-10-CM History of coronary artery 4.4.1 disease I20.89 DX Other forms of angina pectoris ICD-10-CM History of coronary artery 4.4.1 disease I20.1 DX ANGINA PECTORIS WITH DOCUMENTED SPASM ICD-10-CM History of coronary artery 4.4.1 disease I20.8 DX OTHER FORMS OF ANGINA PECTORIS ICD-10-CM History of coronary artery 4.4.1 disease I20.9 DX ANGINA PECTORIS, UNSPECIFIED ICD-10-CM History of coronary artery 4.4.1 disease I20.9 DX ATHEROSCLEROTIC HEART DISEASE OF NATIVE CORONARY ARTERY ATHEROSCLEROTIC HEART DISEASE OF NATIVE CORONARY ARTERY History of coronary artery | | History of coronary artery | | | | |
| 4.4.1 disease History of coronary artery 4.4.1 disease I20.89 DX Other forms of angina pectoris History of coronary artery 4.4.1 disease I20.89 DX Other forms of angina pectoris History of coronary artery 4.4.1 disease I20.1 DX ANGINA PECTORIS WITH DOCUMENTED SPASM History of coronary artery | ICD-10-CM | 4.4.1 disease History of coronary artery IZO.89 DX Angina pectoris with coronary microvascular dysfunction History of coronary artery ICD-10-CM Of the forms of angina pectoris < | | | 120.2 | DX | Refractory angina pectoris | ICD-10-CM |
| 4.4.1 disease I20.89 DX Other forms of angina pectoris History of coronary artery 4.4.1 disease I20.1 DX ANGINA PECTORIS WITH DOCUMENTED SPASM History of coronary artery | | 4.4.1 disease I20.89 DX Other forms of angina pectoris ICD-10-CM History of coronary artery 4.4.1 disease I20.1 DX ANGINA PECTORIS WITH DOCUMENTED SPASM ICD-10-CM 4.4.1 disease I20.8 DX OTHER FORMS OF ANGINA PECTORIS ICD-10-CM History of coronary artery 4.4.1 disease I20.9 DX ANGINA PECTORIS, UNSPECIFIED ICD-10-CM History of coronary artery ATHEROSCLEROTIC HEART DISEASE OF NATIVE CORONARY ARTERY 4.4.1 disease I25.111 DX WITH ANGINA PECTORIS WITH DOCUMENTED SPASM ICD-10-CM History of coronary artery ATHEROSCLEROTIC HEART DISEASE OF NATIVE CORONARY ARTERY | | | 120.81 | DX | Angina pectoris with coronary microvascular dysfunction | ICD-10-CM |
| History of coronary artery 4.4.1 disease I20.1 DX ANGINA PECTORIS WITH DOCUMENTED SPASM History of coronary artery | | History of coronary artery 4.4.1 disease I20.1 DX ANGINA PECTORIS WITH DOCUMENTED SPASM ICD-10-CM History of coronary artery 4.4.1 disease I20.8 DX OTHER FORMS OF ANGINA PECTORIS ICD-10-CM History of coronary artery 4.4.1 disease I20.9 DX ANGINA PECTORIS, UNSPECIFIED ICD-10-CM History of coronary artery 4.4.1 disease I20.9 DX ANGINA PECTORIS, UNSPECIFIED ICD-10-CM ATHEROSCLEROTIC HEART DISEASE OF NATIVE CORONARY ARTERY 4.4.1 disease I25.111 DX WITH ANGINA PECTORIS WITH DOCUMENTED SPASM ICD-10-CM History of coronary artery 4.4.1 disease I25.111 DX ATHEROSCLEROTIC HEART DISEASE OF NATIVE CORONARY ARTERY | | | 120.89 | DX | Other forms of angina pectoris | ICD-10-CM |
| History of coronary artery | ASM ICD-10-CM | History of coronary artery 4.4.1 disease History of coronary artery 4.4.1 disease I20.8 DX OTHER FORMS OF ANGINA PECTORIS ICD-10-CM History of coronary artery 4.4.1 disease I20.9 DX ANGINA PECTORIS, UNSPECIFIED ICD-10-CM ATHEROSCLEROTIC HEART DISEASE OF NATIVE CORONARY ARTERY 4.4.1 disease I25.111 DX WITH ANGINA PECTORIS WITH DOCUMENTED SPASM ICD-10-CM ATHEROSCLEROTIC HEART DISEASE OF NATIVE CORONARY ARTERY 4.4.1 disease I25.111 DX ATHEROSCLEROTIC HEART DISEASE OF NATIVE CORONARY ARTERY | | | | | | |
| | | 4.4.1 disease<br>History of coronary artery IZO.8 DX OTHER FORMS OF ANGINA PECTORIS ICD-10-CM 4.4.1 disease<br>History of coronary artery IZO.9 DX ANGINA PECTORIS, UNSPECIFIED<br>ATHEROSCLEROTIC HEART DISEASE OF NATIVE CORONARY ARTERY ICD-10-CM 4.4.1 disease<br>History of coronary artery IZD.11 DX WITH ANGINA PECTORIS WITH DOCUMENTED SPASM<br>ATHEROSCLEROTIC HEART DISEASE OF NATIVE CORONARY ARTERY ICD-10-CM | | | 120.1 | DX | ANGINA PECTORIS WITH DOCUMENTED SPASM | ICD-10-CM |
| | ICD-10-CM | 4.4.1 disease I20.9 DX ANGINA PECTORIS, UNSPECIFIED ICD-10-CM History of coronary artery ATHEROSCLEROTIC HEART DISEASE OF NATIVE CORONARY ARTERY 4.4.1 disease I25.111 DX WITH ANGINA PECTORIS WITH DOCUMENTED SPASM ATHEROSCLEROTIC HEART DISEASE OF NATIVE CORONARY ARTERY History of coronary artery ATHEROSCLEROTIC HEART DISEASE OF NATIVE CORONARY ARTERY | 4.4.1 | disease | 120.8 | DX | OTHER FORMS OF ANGINA PECTORIS | ICD-10-CM |
| | ICD-10-CM | History of coronary artery 4.4.1 disease I25.111 DX WITH ANGINA PECTORIS WITH DOCUMENTED SPASM ICD-10-CM History of coronary artery ATHEROSCLEROTIC HEART DISEASE OF NATIVE CORONARY ARTERY | | | 120.9 | DX | ANGINA PECTORIS, UNSPECIFIED | ICD-10-CM |
| History of coronary artery ATHEROSCLEROTIC HEART DISEASE OF NATIVE CORONARY ARTER | ATIVE CORONARY ARTERY | History of coronary artery ATHEROSCLEROTIC HEART DISEASE OF NATIVE CORONARY ARTERY | | History of coronary artery | | | ATHEROSCLEROTIC HEART DISEASE OF NATIVE CORONARY ARTERY | |
| | | | | | 125.111 | DX | | ICD-10-CM |
| HISTORY OT CORONARY ARTERY AT HERUSCLERUTIC HEART DISEASE OF NATIVE CURUNARY ARTERY | | | | | 125.118 | DX | WITH OTHER FORMS OF ANGINA PECTORIS | ICD-10-CM |


Componen


BYPASS CORONARY ARTERY, ONE ARTERY FROM LEFT INTERNAL MAMMARY WITH NONAUTOLOGOUS TISSUE


BYPASS INNOMINATE ARTERY TO RIGHT EXTRACRANIAL ARTERY WITH AUTOLOGOUS ARTERIAL TISSUE, OPEN


BYPASS RIGHT SUBCLAVIAN ARTERY TO LEFT LOWER LEG ARTERY WITH NONAUTOLOGOUS TISSUE


BYPASS RIGHT INTERNAL ILIAC ARTERY TO LEFT FEMORAL ARTERY WITH SYNTHETIC SUBSTITUTE,


BYPASS LEFT FEMORAL ARTERY TO LOWER EXTREMITY VEIN WITH NONAUTOLOGOUS TISSUE SUBSTITUTE,


BYPASS LEFT PERONEAL ARTERY TO LOWER EXTREMITY ARTERY WITH AUTOLOGOUS ARTERIAL TISSUE,


OCCLUSION OF LEFT ANTERIOR TIBIAL ARTERY WITH INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC


CONTINUING PREGNANCY AFTER SPONTANEOUS ABORTION OF ONE FETUS OR MORE, SECOND TRIMESTER,


CONTINUING PREGNANCY AFTER INTRAUTERINE DEATH OF ONE FETUS OR MORE, SECOND TRIMESTER, FETUS


CONTINUING PREGNANCY AFTER ELECTIVE FETAL REDUCTION OF ONE FETUS OR MORE, SECOND TRIMESTER,


CEREBRAL INFARCTION DUE TO THROMBOSIS


CEREBRAL INFARCTION DUE TO UNSPECIFIED


MACE component (death, nonfatal MI, nonfatal stroke)


In combination with intravenous administration

In combination with intravenous administration In combination with generic drug name codes for furosemide,

torsemide, bumetanide


AMOXICILLIN, WITH OR WITHOUT


#### Appendix 3. Flowchart for cohort assembly

| OPTUM (Jan 1, 2018 to Feb 28, 2025) | | |
|---|---|---|
| | Excluded Patients | Remaining Patients |
| Patients in dataset | | 95,349,410 |
| Patients meeting cohort entry criteria | | 1,141,594 |
| Excluded due to insufficient enrollment | -375,403 (33%) | 766,191 |
| Excluded due to prior use of referent | -181,012 (24%) | 585,179 |
| Excluded due to prior use of exposure | -292,357 (50%) | 292,822 |
| Excluded because patient qualified in >1 exposure category | -25 (<1%) | 292,797 |
| Excluded based on 1 - Age | -82 (<1%) | 292,715 |
| Excluded based on 1 - Gender | -15 (<1%) | 292,700 |
| Excluded based on 2 - Type 2 diabetes mellitus | -17,966 (6%) | 274,734 |
| Excluded based on 3 - BMI = 25kg/m2 (ICD-10) | -34,519 (13%) | 240,215 |
| Excluded based on 3 - BMI = 25kg/m2 (Truncated) | -879 (<1%) | 239,336 |
| Excluded based on 4 - Increased cardiovascular risk | -3,046 (1%) | 236,290 |
| Excluded based on 5 - History of TIDM or secondary diabetes | -3,008 (1%) | 233,282 |
| Excluded based on 6 - Family or personal history of multiple endocrine neoplasia or medullary thyroid c | -375 (<1%) | 232,907 |
| Excluded based on 7 - End-stage renal disease or dialysis | -1,395 (<1%) | 231,512 |
| Excluded based on 8 - History of treatment for diabetic retinopathy and/or macular edema | -1,700 (<1%) | 229,812 |
| Excluded based on 9 - History of any malignancy | -8,264 (4%) | 221,548 |
| Excluded based on 10 - Cardiovascular event or intervention in the past 7 days | -255 (<1%) | 221,293 |
| Excluded based on 11 - Women who are pregnant or breastfeeding | -101 (<1%) | 221,192 |
| Excluded based on 12 - GLP-1-RA or DPP4i treatment within past 6 months | -8,095 (4%) | 213,097 |
| Excluded based on 13 - Bariatric surgery within the past 12 months | -645 (<1%) | 212,452 |
| Patients in Exposure Group | | 146,733 |
| Patients in Referent Group | | 65,719 |
| Total Patients | | 212.452 |

| MARKETSCAN (Jan 1, 2018 to Dec 31, 2023) | | |
|---|---|---|
| | Excluded Patients | Remaining Patients |
| Patients in dataset | | 126,118,01 |
| Patients meeting cohort entry criteria | | 1,022,94 |
| Excluded due to insufficient enrollment | -213,437 (21%) | 809,50 |
| Excluded due to prior use of referent | -211,348 (26%) | 598,150 |
| Excluded due to prior use of exposure | -345,794 (58%) | 252,36 |
| Excluded because patient qualified in >1 exposure category | -32 (<1%) | 252,33. |
| Excluded based on 1 - Age | -267 (<1%) | 252,06 |
| Excluded based on 1 - Gender | -0 (<1%) | 252,06 |
| Excluded based on 2 - Type 2 diabetes mellitus | -41,509 (16%) | 210,55 |
| Excluded based on 3 - BMI ± 25kg/m2 (ICD-10) | -28,972 (14%) | 181,58: |
| Excluded based on 4 - Increased cardiovascular risk | -4,922 (3%) | 176,66 |
| Excluded based on 5 - History of TIDM or secondary diabetes | -1,941 (1%) | 174,72 |
| Excluded based on 6 - Family or personal history of multiple endocrine neoplasia or meduliary th | -288 (<1%) | 174,43 |
| Excluded based on 7 - End-stage renal disease or dialysis | -479 (<1%) | 173,95 |
| Excluded based on B - History of treatment for diabetic retinopathy and/or macular edema | -682 (<1%) | 173,27 |
| Excluded based on 9 - History of any malignancy | -3,819 (2%) | 169,45 |
| Excluded based on 10 - Cardiovascular event or intervention in the past 7 days | -154 (<1%) | 169,30 |
| Excluded based on 11 - Women who are pregnant or breastfeeding | -172 (<1%) | 169,12 |
| Excluded based on 12 - GLP-1-RA or DPP4i treatment within past 6 months | -5,200 (3%) | 163,92 |
| Excluded based on 13 - Bariatric surgery within the past 12 months | -353 (<1%) | 163,57 |
| Patients in Exposure Group | | 100,97 |
| Patients in Referent Group | | 62,60 |
| Total Patients | | 163.57 |

| MEDICARE (Jan 1, 2018 to Dec 31, 2020) | | |
|---|---|---|
| | Excluded Patients | Remaining Patients |
| Patients in dataset | | 28,874,258 |
| Patients meeting cohort entry criteria | | 953,493 |
| Excluded due to insufficient enrollment | -188,867 (20%) | 764,626 |
| Excluded due to prior use of referent | -551,412 (72%) | 213,214 |
| Excluded due to prior use of exposure | -58,981 (28%) | 154,233 |
| Excluded because patient qualified in >1 exposure category | -17 (<1%) | 154,216 |
| Excluded based on 1 - Age | -0 (<1%) | 154,216 |
| Excluded based on 1 - Gender | -0 (<1%) | 154,216 |
| Excluded based on 2 - Type 2 diabetes mellitus | -2,383 (2%) | 151,833 |
| Excluded based on 3 - BMI ± 25kg/m2 (ICD-10) | -59,852 (39%) | 91,981 |
| Excluded based on 4 - Increased cardiovascular risk | -499 (<1%) | 91,482 |
| Excluded based on 5 - History of TIDM or secondary diabetes | -1,721 (2%) | 89,761 |
| Excluded based on 6 - Family or personal history of multiple endocrine neoplasia or medullary thyroid carcinoma | -168 (<1%) | 89,593 |
| Excluded based on 7 - End-stage renal disease or dialysis | -1,020 (1%) | 88,573 |
| Excluded based on 8 - History of treatment for diabetic retinopathy and/or macular edema | -1,005 (1%) | 87,568 |
| Excluded based on 9 - History of any malignancy | -5,692 (7%) | 81,876 |
| Excluded based on 10 - Cardiovascular event or intervention in the past 7 days | -345 (<1%) | 81,531 |
| Excluded based on 11 - Women who are pregnant or breastfeeding | -6 (<1%) | 81,525 |
| Excluded based on 12 - GLP-1-RA treatment (execpt sema) within past 6 months and DPP4i | -2,959 (4%) | 78,566 |
| Excluded based on 13 - Bariatric surgery within the past 12 months | -257(<1%) | 78,309 |
| Patients in Exposure Group | | 14,653 |
| Patients in Referent Group | | 63,656 |
| Total Patients | | 78,309 |

## Appendix 4.1st Feasibility Assessment

#### Table of Contents

A. Patient characteristics by treatment group B. Summary Parameters of Study Population

C. Median Follow up Time in Overall Study Population
D. Reasons for Censoring in Overall Study Population

E. Initial Power Assessment

F. Aetion report link

G. Review by Principal Investigator

In order to complete the initial power analysis, a dummy outcome of a 90-day gap in database enrollment was used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. We completed a PS overlap weighted comparative analysis using this outcome. The PS included only 3 covariates: age, sex, and combined comorbidity index. Power calculations are based on the formulas from Chow et al. (2008).

OPTUM: Study period from May 13, 2022 to Feb 28, 2025 MARKETSCAN: Study period from May 13, 2022 to Dec 31, 2023

## A. Patient characteristics by treatment group (follow-up start is 1 days after CED, so few patients and dropped, hence table 1 could include sightly fewer patients than the attrition table)

| Before matching | | Optum | | | Marketscan | | | MEDICARE | |
|---|---|---|---|---|---|---|---|---|---|
| Variable | Reference: Sitagliptin | Exposure: Semaglutide injection | Difference | Reference: Sitagliptin | Exposure: Semaglutide injection | Difference | Reference: Sitagliptin | Exposure: Semaglutide injection | Difference |
| Number of patients | 65,719 | 146,733 | - (-, -) | 62,601 | 100,974 | - (-, -) | 63,656 | 14,653 | - (-, -) |
| Age | | | | | | | | | |
| mean (sd) | 69.58 (9.37) | 62.35 (11.30) | 7.23 (7.14, 7.32) | 57.85 (11.73) | 53.66 (9.98) | 4.19 (4.08, 4.30) | 74.01 (6.33) | 71.51 (4.77) | 2.49 (2.40, 2.58) |
| median [IQR] | 70.00 [66.00, 76.00] | 65.00 [55.00, 70.00] | - (-, -) | 58.00 [50.00, 64.00] | 54.00 [47.00, 60.00] | - (-, -) | 73.00 [69.00, 78.00] | 71.00 [68.00, 74.00] | - (-, -) |
| Gender | | | | | | | | | |
| Male; n (%) | 29,191 (44.4%) | 64,543 (44.0%) | 0.4% (-0.0%, 0.9%) | 32,744 (52.3%) | 45,483 (45.0%) | 7.3% (6.8%, 7.8%) | 26,612 (41.8%) | 6,780 (46.3%) | -4.5% (-5.4%, -3.6%) |
| CCI (365 days) | | | | | | | | | |
| mean (sd) | 2.63 (2.78) | 1.96 (2.38) | 0.66 (0.64, 0.69) | 1.14 (1.93) | 1.00 (1.66) | 0.14 (0.12, 0.16) | 2.91 (2.96) | 2.66 (2.59) | 0.24 (0.19, 0.29) |
| median [IQR] | 2.00 [1.00, 4.00] | 1.00 [0.00, 3.00] | - (-, -) | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | - (-, -) | 2.00 [1.00, 5.00] | 2.00 [1.00, 4.00] | - (-, -) |

## B. Summary Parameters of Overall Study Population (Step 1)

| | Optum | Marketscan | MEDICARE |
|---|---|---|---|
| Variable | Value | Value | Value |
| Number of patients in full cohort | 212,452 | 163,575 | 78,309 |
| Number of patients dropped as incomplete cases | 0 | 0 | 0 |
| Number of patients that did not begin follow-up | 403 | 246 | 480 |
| Number of patients in analytic cohort | 212,049 | 163,329 | 77,829 |
| Number of events | 2,976 | 995.00 | 2,743.00 |
| Number of person-years | 111,210.65 | 87,462.82 | 40,508.35 |
| Number of patients in group: Reference- Sitagliptin | 65,509 | 62,460 | 63,194 |
| Number of patients in group: Exposure - Tirzepatide | 146,540 | 100,869 | 14,635 |
| Risk per 1,000 patients | 14.03 | 6.09 | 35.24 |
| Rate per 1,000 person-years | 26.76 | 11.38 | 67.71 |

# C. Median Follow up Time in Overall Study Population (Step 1)

| | Optum | Marketscan | MEDICARE |
|---|---|---|---|
| Patient Group | Median Follow-Up | Median Follow-Up Time | Median Follow-Up |
| Overall Patient Population | 159 [92, 309] | 166 [88, 325] | 153 [84, 313] |

# D. Reasons for Censoring in Overall Study Population (Step 1)

| | Optum | Marketscan | MEDICARE |
|---|---|---|---|
| Overall | Value | Value | Value |
| Outcome | 2,976 (1.4%) | 995 (0.6%) | 2,743 (3.5%) |
| Start of an additional exposure | 1,949 (0.9%) | 2,484 (1.5%) | 652 (0.8%) |
| End of index exposure | 99,298 (46.8%) | 66,775 (40.9%) | 33,724 (43.3%) |
| Maximum follow-up time | 42,557 (20.1%) | 35,381 (21.7%) | 15,361 (19.7%) |
| Specified date reached | 7,745 (3.7%) | 28,075 (17.2%) | 13,789 (17.7%) |
| End of patient data | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) |
| End of patient enrollment | 42,381 (20.0%) | 19,063 (11.7%) | 2,959 (3.8%) |
| Switch to other GLP-1-RA (for censoring) / Nursing home admission | 15,143 (7.1%) | 10,556 (6.5%) | 8,601 (11.1%) |

# E. Power Assessment

| Superiority Analysis | Optum | Marketscan | Medicare |
|---------------------------|---------|------------|----------|
| Number of patients | | | |
| Reference | 65,719 | 62,601 | 63,656 |
| Exposed | 146,733 | 100,974 | 14,653 |
| Risk per 1,000 patients | 14.03 | 6.09 | 35.24 |
| Expected HR | 0.7 | 0.7 | 0.7 |
| Alpha (2-sided) | 0.05 | 0.05 | 0.05 |
| Number of events expected | 2981 | 996 | 2760 |

| Power | 1.00 | 1.00 | 1.00 |
|-------|------|------|------|

F. Aetion report link
Ontum Step 1: https://hwh-dope.aetion.com/project/2914/rwrs/139463
Marketscan Step 1: https://bwh-dope.aetion.com/project/2912/rwrs/139471
Medicare Step 1: https://bwh-dope.aetion.com/project/2913/rwrs/139471

# F. Review by principal investigator

Stop analyses until feasibility and power are reviewed by primary investigators.

| Reviewed by PI: | Nils Krüger | Date reviewed: | July 30, 202 |
|-----------------|-------------|----------------|--------------|

#### Appendix 5. 2nd Feasibility Assessment

## Table of Contents

A. Median Follow up Time by Treatment Group B. Reasons for Censoring by Treatment Group C. Final Power Assessment D. Aetion report link E. Review by Principal Investigator

In order to complete the feasibility analysis, a dummy outcome of a 90-day gap in database enrollment was used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. We completed a PS overlap weighted comparative analysis using this outcome. The PS included all prespecified covariates listed in the protocol. Power calculations are based on the formulas from Chow et al. (2008).

## A. Median Follow Up Time by Treatment Group

| | Median Follow-Up | Median Follow-Up Time (Days) | Median Follow-Up Time (Days) |
|---|---|---|---|
| Patient Group | Time (Days) [IQR] | [IQR] | [IQR] |
| Overall Patient Population | 159 [92, 309] | 166 [88, 325] | 153 [84, 313] |

## B. Reasons for Censoring in Overall Study Population

| | Optum | Marketscan | MEDICARE |
|---|---|---|---|
| Overall | Value | Value | Value |
| Outcome | 2,976 (1.4%) | 995 (0.6%) | 2,743 (3.5%) |
| Start of an additional exposure | 1,949 (0.9%) | 2,484 (1.5%) | 652 (0.8%) |
| End of index exposure | 99,298 (46.8%) | 66,775 (40.9%) | 33,724 (43.3%) |
| Maximum follow-up time | 42,557 (20.1%) | 35,381 (21.7%) | 15,361 (19.7%) |
| Specified date reached | 7,745 (3.7%) | 28,075 (17.2%) | 13,789 (17.7%) |
| End of patient data | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) |
| End of patient enrollment | 42,381 (20.0%) | 19,063 (11.7%) | 2,959 (3.8%) |
| Switch to other GLP-1-RA (for censoring) / Nursing home admission | 15,143 (7.1%) | 10,556 (6.5%) | 8,601 (11.1%) |

## C. Power Assessment

| Superiority Analysis | Optum | Marketscan | Medicare |
|---------------------------|---------|------------|----------|
| Number of patients | | | |
| Reference | 65,719 | 62,601 | 63,656 |
| Exposed | 146,733 | 100,974 | 14,653 |
| Risk per 1,000 patients | 14.03 | 6.09 | 35.24 |
| Expected HR | 0.7 | 0.7 | 0.7 |
| Alpha (2-sided) | 0.05 | 0.05 | 0.05 |
| Number of events expected | 2981 | 996 | 2760 |
| Power | 1.00 | 1.00 | 1.00 |

#### D. Aetion report link

Optum Step 1: https://bwh-dopeaetion.com/project/2914/rwrs/139463
Marketscan Step 1: https://bwh-dopeaetion.com/project/2912/rwrs/139471
Medicare Step 1: https://bwh-dopeaetion.com/project/2913/rwrs/139477

# E. Review by principal investigator

Stop analyses until feasibility and power are reviewed by primary investigators.

| Reviewed by PI: | Nils Krüger | Date reviewed: | July 30, 2025 |
|-----------------|-------------|----------------|---------------|

## Appendix 6. Balance Assessment - PS Distribution and C-Statistic

## C-statistics unadjusted, OPTUM: 0.888



#### C-statistics adjusted after overlap weighing on the PS, OPTUM: 0.518



## C-statistics unadjusted, MARKETSCAN: 0.864



C-statistics adjusted after overlap weighing on the PS, MARKETSCAN: 0.520



## C-statistics unadjusted, MEDICARE: 0.836



#### C-statistics adjusted after overlap weighing on the PS, MEDICARE: 0.524



Appendix 7. Balance Assessment - Table 1

| ОРТИМ | | | | | | |
|---|---|---|---|---|---|---|
| Variable | Reference: Sitagliptin | Exposure: Semaglutide injection | Difference | Reference: Sitagliptin | Exposure: Semaglutide injection | Difference |
| Number of patients | 65,509 | 146,540 | - (-, -) | 33.973 | 33,973 | - (-, -) |
| Year of Cohort Entry Date | 03,303 | 140,540 | - (-, -) | 33,373 | 33,373 | - (-, -) |
| 2018; n (%) | 12,168 (18.6%) | 193 (0.1%) | 18.4% (18.1%, 18.7%) | 217 (0.6%) | 193 (0.6%) | 0.1% (-0.0%, 0.2%) |
| 2019; n (%) | 11,876 (18.1%) | 5,785 (3.9%) | 14.2% (13.9%, 14.5%) | 3,836 (11.3%) | 3,962 (11.7%) | -0.4% (-0.9%, 0.1%) |
| 2015, II (70)<br>2020; n (%) | 10,642 (16.2%) | 8,825 (6.0%) | 10.2% (9.9%, 10.5%) | 4,986 (14.7%) | 5,033 (14.8%) | -0.1% (-0.7%, 0.4%) |
| 2021; n (%) | 9,335 (14.2%) | 14,639 (10.0%) | 4.3% (4.0%, 4.6%) | 5,898 (17.4%) | 5,951 (17.5%) | -0.1% (-0.7%, 0.4%) |
| 2021; n (%) | 7.776 (11.9%) | 24,189 (16.5%) | -4.6% (-4.9%, -4.3%) | 6,275 (18.5%) | 6.202 (18.3%) | 0.2% (-0.4%, 0.8%) |
| 2023; n (%) | 6,935 (10.6%) | 44.241 (30.2%) | -19.6% (-19.9%, -19.3%) | 6,275 (18.5%) | 6,366 (18,7%) | 0.1% (-0.5%, 0.7%) |
| | 6,742 (10.3%) | 47,352 (32.3%) | -19.6% (-19.9%, -19.5%) | 6,323 (18.6%) | 6,225 (18.3%) | 0.3% (-0.3%, 0.7%) |
| 2024; n (%)<br>2025; n (%) | 35 (0.1%) | 1,316 (0.9%) | -0.8% (-0.9%, -0.8%) | | | -0.0% (-0.1%, 0.0%) |
| | 35 (0.1%) | 1,316 (0.9%) | -0.8% (-0.9%, -0.8%) | 33 (0.1%) | 41 (0.1%) | -0.0% (-0.1%, 0.0%) |
| Age | CO E7 (0.26) | C2 25 (11 20) | 7.02 (7.14 7.20) | 67.00 (0.61) | C7 70 (0.22) | 0.11 ( 0.02 (0.05) |
| mean (sd) | 69.57 (9.36) | 62.35 (11.30) | 7.23 (7.14, 7.32) | 67.89 (9.61) | 67.78 (9.32) | 0.11 (-0.03, 0.25) |
| median [IQR] | 70.00 [66.00, 76.00] | 65.00 [55.00, 70.00] | - (-, -) | 69.00 [64.00, 74.00] | 69.00 [63.00, 74.00] | - (-, -) |
| min, max | 20.00, 88.00 | 18.00, 88.00 | - (-, -) | 20.00, 88.00 | 25.00, 88.00 | - (-, -) |
| Gender (male); n (%) | 29,099 (44.4%) | 64,467 (44.0%) | 0.4% (-0.0%, 0.9%) | 14,946 (44.0%) | 14,960 (44.0%) | -0.0% (-0.8%, 0.7%) |
| Race (Recategorized) | <b></b> | | | | | |
| White; n (%) | 28,948 (44.2%) | 66,030 (45.1%) | -0.9% (-1.3%, -0.4%) | 15,554 (45.8%) | 15,545 (45.8%) | 0.0% (-0.7%, 0.8%) |
| Black; n (%) | 11,899 (18.2%) | 19,891 (13.6%) | 4.6% (4.2%, 4.9%) | 5,684 (16.7%) | 5,757 (16.9%) | -0.2% (-0.8%, 0.4%) |
| Unknown / Missing; n (%) | 22,514 (34.4%) | 58,262 (39.8%) | -5.4% (-5.8%, -4.9%) | 11,962 (35.2%) | 11,895 (35.0%) | 0.2% (-0.5%, 0.9%) |
| Others; n (%) | 2,148 (3.3%) | 2,357 (1.6%) | 1.7% (1.5%, 1.8%) | 773 (2.3%) | 776 (2.3%) | -0.0% (-0.2%, 0.2%) |
| Region / State | | | | | | |
| Northest; n (%) | 7,242 (11.1%) | 12,799 (8.7%) | 2.3% (2.0%, 2.6%) | 3,605 (10.6%) | 3,569 (10.5%) | 0.1% (-0.4%, 0.6%) |
| Midwest / North central; n (%) | 9,310 (14.2%) | 30,398 (20.7%) | -6.5% (-6.9%, -6.2%) | 5,673 (16.7%) | 5,604 (16.5%) | 0.2% (-0.4%, 0.8%) |
| South; n (%) | 37,213 (56.8%) | 80,054 (54.6%) | 2.2% (1.7%, 2.6%) | 19,073 (56.1%) | 19,152 (56.4%) | -0.2% (-1.0%, 0.5%) |
| West; n (%) | 11,710 (17.9%) | 23,230 (15.9%) | 2.0% (1.7%, 2.4%) | 5,608 (16.5%) | 5,632 (16.6%) | -0.1% (-0.6%, 0.5%) |
| Missing; n (%) | 34 (0.1%) | 59 (0.0%) | 0.0% (-0.0%, 0.0%) | 14 (0.0%) | 16 (0.0%) | -0.0% (-0.0%, 0.0%) |
| Smoking/Tobacco use; n (%) | 16,044 (24.5%) | 35,849 (24.5%) | 0.0% (-0.4%, 0.4%) | 8,376 (24.7%) | 8,395 (24.7%) | -0.1% (-0.7%, 0.6%) |
| Weight | | | | | | |
| Underweight; n (%) | 64 (0.1%) | 41 (0.0%) | 0.1% (0.0%, 0.1%) | 13 (0.0%) | 15 (0.0%) | -0.0% (-0.0%, 0.0%) |
| Normal weight; n (%) | 1,170 (1.8%) | 424 (0.3%) | 1.5% (1.4%, 1.6%) | 280 (0.8%) | 270 (0.8%) | 0.0% (-0.1%, 0.2%) |
| Overweight; n (%) | 17,125 (26.1%) | 15,116 (10.3%) | 15.8% (15.5%, 16.2%) | 6,744 (19.9%) | 6,789 (20.0%) | -0.1% (-0.7%, 0.5%) |
| Class 1 Obesity; n (%) | 10,018 (15.3%) | 14,784 (10.1%) | 5.2% (4.9%, 5.5%) | 4,756 (14.0%) | 4,777 (14.1%) | -0.1% (-0.6%, 0.5%) |
| Class 2 Obesity; n (%) | 4,424 (6.8%) | 10,306 (7.0%) | -0.3% (-0.5%, -0.0%) | 2,439 (7.2%) | 2,409 (7.1%) | 0.1% (-0.3%, 0.5%) |
| Class 3 Obesity; n (%) | 14,046 (21.4%) | 58,436 (39.9%) | -18.4% (-18.8%, -18.0%) | 9,206 (27.1%) | 9,132 (26.9%) | 0.2% (-0.5%, 0.9%) |
| Unspecified Obesity; n (%) | 18,662 (28.5%) | 47,433 (32.4%) | -3.9% (-4.3%, -3.5%) | 10,535 (31.0%) | 10,581 (31.1%) | -0.1% (-0.8%, 0.6%) |
| Diabetic retinopathy; n (%) | 7,021 (10.7%) | 12,474 (8.5%) | 2.2% (1.9%, 2.5%) | 3,457 (10.2%) | 3,514 (10.3%) | -0.2% (-0.6%, 0.3%) |
| Diabetic neuropathy; n (%) | 21,697 (33.1%) | 38,182 (26.1%) | 7.1% (6.6%, 7.5%) | 10,697 (31.5%) | 10,890 (32.1%) | -0.6% (-1.3%, 0.1%) |
| Diabetic nephropathy; n (%) | 19,291 (29.4%) | 30,714 (21.0%) | 8.5% (8.1%, 8.9%) | 9,049 (26.6%) | 9,148 (26.9%) | -0.3% (-1.0%, 0.4%) |
| Diabetes with other ophthalmic complications; n (%) | 4,010 (6.1%) | 5,844 (4.0%) | 2.1% (1.9%, 2.3%) | 1,886 (5.6%) | 1,948 (5.7%) | -0.2% (-0.5%, 0.2%) |
| Diabetes with peripheral circulatory disorders; n (%) | 11,814 (18.0%) | 20,462 (14.0%) | 4.1% (3.7%, 4.4%) | 5,882 (17.3%) | 5,878 (17.3%) | 0.0% (-0.6%, 0.6%) |
| Diabetic foot; n (%) | 2,161 (3.3%) | 4,359 (3.0%) | 0.3% (0.2%, 0.5%) | 1,088 (3.2%) | 1,123 (3.3%) | -0.1% (-0.4%, 0.2%) |
| Erectile dysfunction; n (%) | 2,631 (4.0%) | 7,345 (5.0%) | -1.0% (-1.2%, -0.8%) | 1,492 (4.4%) | 1,531 (4.5%) | -0.1% (-0.4%, 0.2%) |
| Hypoglycemia; n (%) | 16,711 (25.5%) | 35,046 (23.9%) | 1.6% (1.2%, 2.0%) | 8,722 (25.7%) | 8,717 (25.7%) | 0.0% (-0.6%, 0.7%) |
| Hyperglycemia/DKA/HONK; n (%) | 34,625 (52.9%) | 75,069 (51.2%) | 1.6% (1.2%, 2.1%) | 18,004 (53.0%) | 18,118 (53.3%) | -0.3% (-1.1%, 0.4%) |
| Skin infections; n (%) | 6,799 (10.4%) | 15,469 (10.6%) | -0.2% (-0.5%, 0.1%) | 3,544 (10.4%) | 3,601 (10.6%) | -0.2% (-0.6%, 0.3%) |
| Stable angina; n (%) | 3,404 (5.2%) | 7,012 (4.8%) | 0.4% (0.2%, 0.6%) | 1,718 (5.1%) | 1,758 (5.2%) | -0.1% (-0.5%, 0.2%) |
| Unstable angina; n (%) | 1,961 (3.0%) | 3,596 (2,5%) | 0.5% (0.4%, 0.7%) | 926 (2.7%) | 943 (2.8%) | -0.1% (-0.3%, 0.2%) |
| Hypertension; n (%) | 60,446 (92.3%) | 129,348 (88.3%) | 4.0% (3.7%, 4.3%) | 31,001 (91.3%) | 30,983 (91.2%) | 0.1% (-0.4%, 0.5%) |
| Hypotension; n (%) | 2,748 (4.2%) | 4,294 (2.9%) | 1.3% (1.1%, 1.4%) | 1,255 (3.7%) | 1,293 (3.8%) | -0.1% (-0.4%, 0.2%) |
| Hyperlipidemia; n (%) | 57,587 (87.9%) | 124,937 (85.3%) | 2.6% (2.3%, 3.0%) | 29,727 (87.5%) | 29,853 (87.9%) | -0.4% (-0.9%, 0.1%) |
| Atrial fibrillation; n (%) | 7,859 (12.0%) | 14,252 (9.7%) | 2.3% (2.0%, 2.6%) | 3,897 (11.5%) | 3,849 (11.3%) | 0.1% (-0.3%, 0.6%) |
| Cardiac conduction disorder; n (%) | 4,498 (6.9%) | 8,245 (5.6%) | 1.2% (1.0%, 1.5%) | 2,229 (6,6%) | 2,231 (6.6%) | -0.0% (-0.4%, 0.4%) |
| Previous cardiac procedure (CABG, PTCA, Stent); n (%) | 1.178 (1.8%) | 2.505 (1.7%) | 0.1% (-0.0%, 0.2%) | 578 (1.7%) | 621 (1.8%) | -0.1% (-0.3%, 0.1%) |
| Ischemic stroke; n (%) | 719 (1.1%) | 978 (0.7%) | 0.4% (0.3%, 0.5%) | 298 (0.9%) | 313 (0.9%) | -0.0% (-0.2%, 0.1%) |
| PVD diagnosis or surgery; n (%) | 9,099 (13.9%) | 13,697 (9.3%) | 4.5% (4.2%, 4.8%) | 4,208 (12.4%) | 4,271 (12.6%) | -0.2% (-0.7%, 0.3%) |
| Other cardiac dysrhythmia; n (%) | 14,125 (21.6%) | 29,604 (20.2%) | 1.4% (1.0%, 1.7%) | 7,164 (21.1%) | 7,175 (21.1%) | -0.2% (-0.7%, 0.3%) |
| | 4,004 (6.1%) | 7,488 (5.1%) | 1.0% (0.8%, 1.2%) | 1,919 (5.6%) | 1,877 (5.5%) | 0.1% (-0.2%, 0.5%) |
| Cardiomyopathy; n (%) Valve disorders; n (%) | 8,567 (13.1%) | 7,488 (5.1%)<br>15,354 (10.5%) | 2.6% (2.3%, 2.9%) | 4,202 (12.4%) | 4,186 (12.3%) | 0.1% (-0.2%, 0.5%) |
| | | | | 4,202 (12.4%) | 4,186 (12.3%) | |
| Valve replacement; n (%) | 951 (1.5%) | 1,667 (1.1%) | 0.3% (0.2%, 0.4%) | 1 7 | | 0.0% (-0.2%, 0.2%) |
| TIA; n (%) | 1,592 (2.4%) | 2,479 (1.7%) | 0.7% (0.6%, 0.9%) | 678 (2.0%) | 677 (2.0%) | 0.0% (-0.2%, 0.2%) |
| Edema; n (%) | 9,890 (15.1%) | 20,415 (13.9%) | 1.2% (0.8%, 1.5%) | 5,007 (14.7%) | 5,020 (14.8%) | -0.0% (-0.6%, 0.5%) |

| Venezia there as hadio as / Dulas as a sankalia as a /0/\ | 2,376 (3,6%) | 4.777 (3.3%) | 0.4% (0.2%, 0.5%) | 1,191 (3,5%) | 1.172 (3.4%) | 0.1% (-0.2%, 0.3%) |
|---|---|---|---|---|---|---|
| Venous thromboembolism / Pulmonary embolism; n (%) Pulmonary hypertension; n (%) | 2,449 (3.7%) | 4,393 (3.0%) | 0.4% (0.2%, 0.5%) | 1,191 (3.5%) | 1,172 (3.4%) | 0.1% (-0.2%, 0.3%) |
| Implantable cardioverter defibrillator; n (%) | 239 (0.4%) | 349 (0.2%) | 0.1% (0.1%, 0.2%) | 107 (0.3%) | 103 (0.3%) | 0.0% (-0.1%, 0.1%) |
| Hyperkalemia: n (%) | 2,982 (4.6%) | 4,343 (3.0%) | 1.6% (1.4%, 1.8%) | 1,356 (4.0%) | 1,352 (4.0%) | 0.0% (-0.1%, 0.1%) |
| Coronary atherosclerosis; n (%) | 16,289 (24.9%) | 31,160 (21.3%) | 3.6% (3.2%, 4.0%) | 8.131 (23.9%) | 8,157 (24.0%) | -0.1% (-0.7%, 0.6%) |
| Cerebrovascular procedure; n (%) | 125 (0.2%) | 202 (0.1%) | 0.1% (0.0%, 0.1%) | 59 (0.2%) | 66 (0.2%) | -0.0% (-0.1%, 0.0%) |
| Insertion of pacemakers / removal of cardiac lead; n (%) | 207 (0.3%) | 225 (0.2%) | 0.2% (0.1%, 0.2%) | 78 (0.2%) | 87 (0.3%) | -0.0% (-0.1%, 0.1%) |
| CKD Stage 1-2; n (%) | 5,345 (8.2%) | 7,718 (5.3%) | 2.9% (2.7%, 3.1%) | 2,389 (7.0%) | 2,427 (7.1%) | -0.1% (-0.5%, 0.3%) |
| CKD Stage 3-4; n (%) | 14,299 (21.8%) | 22,030 (15.0%) | 6.8% (6.4%, 7.2%) | 6,729 (19.8%) | 6,744 (19.9%) | -0.0% (-0.6%, 0.6%) |
| Unspecified CKD; n (%) | 5,698 (8.7%) | 8,740 (6.0%) | 2.7% (2.5%, 3.0%) | 2,663 (7.8%) | 2,656 (7.8%) | 0.0% (-0.4%, 0.4%) |
| Acute kidney injury; n (%) | 6,159 (9.4%) | 8,885 (6.1%) | 3.3% (3.1%, 3.6%) | 2,733 (8.0%) | 2,767 (8.1%) | -0.1% (-0.5%, 0.3%) |
| Hypertensive nephropathy; n (%) | 11,888 (18.1%) | 18,427 (12.6%) | 5.6% (5.2%, 5.9%) | 5,562 (16.4%) | 5,615 (16.5%) | -0.2% (-0.7%, 0.4%) |
| Urinary tract infections; n (%) | 11,376 (17.4%) | 19,129 (13.1%) | 4.3% (4.0%, 4.7%) | 5,305 (15.6%) | 5,302 (15.6%) | 0.0% (-0.5%, 0.6%) |
| Genital infections; n (%) | 2,508 (3.8%) | 5,201 (3.5%) | 0.3% (0.1%, 0.5%) | 1,302 (3.8%) | 1,338 (3.9%) | -0.1% (-0.4%, 0.2%) |
| Urolithiasis (Kidney and urinary stone); n (%) | 2,947 (4.5%) | 6,716 (4.6%) | -0.1% (-0.3%, 0.1%) | 1,557 (4.6%) | 1,569 (4.6%) | -0.0% (-0.4%, 0.3%) |
| COPD; n (%) | 10,525 (16.1%) | 18,765 (12.8%) | 3.3% (2.9%, 3.6%) | 5,173 (15.2%) | 5,232 (15.4%) | -0.2% (-0.7%, 0.4%) |
| Asthma; n (%) | 7,158 (10.9%) | 18,901 (12.9%) | -2.0% (-2.3%, -1.7%) | 3,994 (11.8%) | 4,037 (11.9%) | -0.1% (-0.6%, 0.4%) |
| Obstructive sleep apnea; n (%) | 13,320 (20.3%) | 48,510 (33.1%) | -12.8% (-13.2%, -12.4%) | 8,413 (24.8%) | 8,479 (25.0%) | -0.2% (-0.8%, 0.5%) |
| Serious bacterial infections; n (%) | 2,706 (4.1%) | 3,924 (2.7%) | 1.5% (1.3%, 1.6%) | 1,171 (3.4%) | 1,159 (3.4%) | 0.0% (-0.2%, 0.3%) |
| Pneumonia; n (%) | 4,213 (6.4%) | 7,210 (4.9%) | 1.5% (1.3%, 1.7%) | 1,985 (5.8%) | 1,953 (5.7%) | 0.1% (-0.3%, 0.4%) |
| Liver disease; n (%) | 11,081 (16.9%) | 26,199 (17.9%) | -1.0% (-1.3%, -0.6%) | 5,925 (17.4%) | 5,929 (17.5%) | -0.0% (-0.6%, 0.6%) |
| MASH/MASLD; n (%) | 4,960 (7.6%) | 15,221 (10.4%) | -2.8% (-3.1%, -2.6%) | 2,911 (8.6%) | 2,970 (8.7%) | -0.2% (-0.6%, 0.3%) |
| Fractures / Falls; n (%) | 5,129 (7.8%) | 8,413 (5.7%) | 2.1% (1.8%, 2.3%) | 2,459 (7.2%) | 2,455 (7.2%) | 0.0% (-0.4%, 0.4%) |
| Osteoporosis; n (%) | 4,315 (6.6%) | 6,308 (4.3%) | 2.3% (2.1%, 2.5%) | 1,992 (5.9%) | 1,969 (5.8%) | 0.1% (-0.3%, 0.4%) |
| Osteoarthritis; n (%) | 21,532 (32.9%) | 45,336 (30.9%) | 1.9% (1.5%, 2.4%) | 11,097 (32.7%) | 11,056 (32.5%) | 0.1% (-0.6%, 0.8%) |
| Depression; n (%) | 14,524 (22.2%) | 34,185 (23.3%) | -1.2% (-1.5%, -0.8%) | 7.631 (22.5%) | 7.715 (22.7%) | -0.2% (-0.9%, 0.4%) |
| Dementia; n (%) | 4,845 (7.4%) | 4,391 (3.0%) | 4.4% (4.2%, 4.6%) | 1,820 (5.4%) | 1,886 (5.6%) | -0.2% (-0.5%, 0.2%) |
| Delirium or psychosis; n (%) | 1,755 (2.7%) | 2,406 (1.6%) | 1.0% (0.9%, 1.2%) | 761 (2.2%) | 803 (2.4%) | -0.1% (-0.4%, 0.1%) |
| Anxiety; n (%) | 11,583 (17.7%) | 34,402 (23.5%) | -5.8% (-6.2%, -5.4%) | 6,566 (19.3%) | 6,608 (19.5%) | -0.1% (-0.7%, 0.5%) |
| Sleep disorders; n (%) | 23,188 (35.4%) | 53,052 (36.2%) | -0.8% (-1.2%, -0.4%) | 12,067 (35.5%) | 12,209 (35.9%) | -0.4% (-1.1%, 0.3%) |
| Anemia; n (%) | 15,037 (23.0%) | 26,540 (18.1%) | 4.8% (4.5%, 5.2%) | 7,203 (21.2%) | 7,256 (21.4%) | -0.2% (-0.8%, 0.5%) |
| Influenza; n (%) | 1,131 (1.7%) | 2,568 (1.8%) | -0.0% (-0.1%, 0.1%) | 502 (1.5%) | 498 (1.5%) | 0.0% (-0.2%, 0.2%) |
| COVID: n (%) | 3,375 (5.2%) | 14.783 (10.1%) | -4.9% (-5.2%, -4.7%) | 2,593 (7.6%) | 2,480 (7.3%) | 0.3% (-0.1%, 0.7%) |
| Hyperthyroidism and other thyroid gland disorders; n (%) | 17,304 (26.4%) | 38,345 (26.2%) | 0.2% (-0.2%, 0.7%) | 8,954 (26.4%) | 8,996 (26.5%) | -0.1% (-0.8%, 0.5%) |
| Hypothyroidism; n (%) | 14.224 (21.7%) | 31,043 (21.2%) | 0.5% (0.1%, 0.9%) | 7,358 (21.7%) | 7,357 (21.7%) | 0.0% (-0.6%, 0.6%) |
| Nephrotic syndrome; n (%) | 57 (0.1%) | 140 (0.1%) | -0.0% (-0.0%, 0.0%) | 25 (0.1%) | 24 (0.1%) | 0.0% (-0.0%, 0.0%) |
| Urinary incontinence; n (%) | 4,393 (6.7%) | 8,269 (5.6%) | 1.1% (0.8%, 1.3%) | 2,219 (6.5%) | 2,308 (6.8%) | -0.3% (-0.6%, 0.1%) |
| Biliary disease; n (%) | 164 (0.3%)<br>107 (0.2%) | 201 (0.1%)<br>147 (0.1%) | 0.1% (0.1%, 0.2%) | 81 (0.2%)<br>42 (0.1%) | 68 (0.2%)<br>39 (0.1%) | 0.0% (-0.0%, 0.1%) |
| Pancreatitis; n (%) | | | 0.1% (0.0%, 0.1%) | | | 0.0% (-0.0%, 0.1%) |
| Bowel obstruction; n (%) | 99 (0.2%) | 149 (0.1%) | 0.0% (0.0%, 0.1%) | 46 (0.1%) | 47 (0.1%) | -0.0% (-0.1%, 0.1%) |
| Gastroparesis; n (%) | 639 (1.0%) | 1,193 (0.8%) | 0.2% (0.1%, 0.3%) | 344 (1.0%) | 375 (1.1%) | -0.1% (-0.2%, 0.1%) |
| Number of antidiabetic drugs on CED | | | | | | |
| mean (sd) | 2.24 (0.85) | 2.08 (0.90) | 0.16 (0.15, 0.17) | 2.22 (0.87) | 2.24 (0.91) | -0.02 (-0.03, -0.01) |
| median [IQR] | 2.00 [2.00, 3.00] | 2.00 [1.00, 3.00] | - (-, -) | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | - (-, -) |
| min, max | 1.00, 6.00 | 1.00, 6.00 | - (-, -) | 1.00, 6.00 | 1.00, 6.00 | - (-, -) |
| Concomitant use or initiation of Metformin; n (%) | 40,064 (61.2%) | 74,154 (50.6%) | 10.6% (10.1%, 11.0%) | 19,703 (58.0%) | 19,850 (58.4%) | -0.4% (-1.2%, 0.3%) |
| Concomitant use or initiation of Insulins; n (%) | 8,830 (13.5%) | 28,757 (19.6%) | -6.1% (-6.5%, -5.8%) | 5,552 (16.3%) | 5,752 (16.9%) | -0.6% (-1.2%, -0.0%) |
| Concomitant use or initiation of Sulfonylureas; n (%) | 20,225 (30.9%) | 23,766 (16.2%) | 14.7% (14.3%, 15.1%) | 8,739 (25.7%) | 8,839 (26.0%) | -0.3% (-1.0%, 0.4%) |
| Concomitant use or initiation of SGLT-2i; n (%) | 6,999 (10.7%) | 23,236 (15.9%) | -5.2% (-5.5%, -4.9%) | 4,884 (14.4%) | 5,063 (14.9%) | -0.5% (-1.1%, 0.0%) |
| Concomitant use or initiation of Any other glucose-lowering drugs; n (%) | 4,817 (7.4%) | 8,009 (5.5%) | 1.9% (1.7%, 2.1%) | 2,424 (7.1%) | 2,458 (7.2%) | -0.1% (-0.5%, 0.3%) |
| Past use of Metformin; n (%) | 46,144 (70.4%) | 97,987 (66.9%) | 3.6% (3.1%, 4.0%) | 23,689 (69.7%) | 23,832 (70.1%) | -0.4% (-1.1%, 0.3%) |
| Past use of Insulins; n (%) | 12,255 (18.7%) | 37,726 (25.7%) | -7.0% (-7.4%, -6.7%) | 7,505 (22.1%) | 7,722 (22.7%) | -0.6% (-1.3%, -0.0%) |
| Past use of Sulfonylureas; n (%) | 26,215 (40.0%) | 33,839 (23.1%) | 16.9% (16.5%, 17.4%) | 11,663 (34.3%) | 11,803 (34.7%) | -0.4% (-1.1%, 0.3%) |
| Past use of SGLT-2i; n (%) | 10,505 (16.0%) | 32,183 (22.0%) | -5.9% (-6.3%, -5.6%) | 7,109 (20.9%) | 7,322 (21.6%) | -0.6% (-1.2%, -0.0%) |
| Past use of Any other glucose-lowering drugs; n (%) | 6,939 (10.6%) | 11,263 (7.7%) | 2.9% (2.6%, 3.2%) | 3,442 (10.1%) | 3,468 (10.2%) | -0.1% (-0.5%, 0.4%) |
| ACE-is/ARB's; n (%) | 51,282 (78.3%) | 106,815 (72.9%) | 5.4% (5.0%, 5.8%) | 26,030 (76.6%) | 26,037 (76.6%) | -0.0% (-0.7%, 0.6%) |
| ARNI; n (%) | 770 (1.2%) | 2,511 (1.7%) | -0.5% (-0.6%, -0.4%) | 486 (1.4%) | 462 (1.4%) | 0.1% (-0.1%, 0.2%) |
| Thiazides; n (%) | 23,234 (35.5%) | 51,553 (35.2%) | 0.3% (-0.2%, 0.7%) | 12,037 (35.4%) | 11,993 (35.3%) | 0.1% (-0.6%, 0.9%) |
| Beta-blockers; n (%) | 31,100 (47.5%) | 61,361 (41.9%) | 5.6% (5.1%, 6.1%) | 15,686 (46.2%) | 15,569 (45.8%) | 0.3% (-0.4%, 1.1%) |
| Calcium channel blockers; n (%) | 24,798 (37.9%) | 47,975 (32.7%) | 5.1% (4.7%, 5.6%) | 12,414 (36.5%) | 12,433 (36.6%) | -0.1% (-0.8%, 0.7%) |
| Digoxin / Digitoxin; n (%) | 818 (1.2%) | 903 (0.6%) | 0.6% (0.5%, 0.7%) | 325 (1.0%) | 323 (1.0%) | 0.0% (-0.1%, 0.2%) |
| Loop diuretics; n (%) | 13,192 (20.1%) | 27,529 (18.8%) | 1.4% (1.0%, 1.7%) | 6,782 (20.0%) | 6,761 (19.9%) | 0.1% (-0.5%, 0.7%) |
| Other diuretics: n (%) | 5.134 (7.8%) | 13.715 (9.4%) | -1.5% (-1.8%, -1.3%) | 2.871 (8.5%) | 2.857 (8.4%) | 0.0% (-0.4%, 0.5%) |
| Intravenous diuretics; n (%) | 1,105 (1.7%) | 2,069 (1.4%) | 0.3% (0.2%, 0.4%) | 536 (1.6%) | 542 (1.6%) | -0.0% (-0.2%, 0.2%) |
| Nitrates; n (%) | 5,044 (7.7%) | 9,447 (6.4%) | 1.3% (1.0%, 1.5%) | | | -0.2% (-0.6%, 0.2%) |
| INIUates, II (70) | 3,044 (7.7%) | J,441 (0.470) | 1.370 (1.U%, 1.3%) | 2,426 (7.1%) | 2,501 (7.4%) | -U.2% (-U.0%, U.2%) |

| A of the Horizon of Mark | 1.631 (2.5%) | 3.413 (2.3%) | 0.2% (0.0%, 0.3%) | 851 (2.5%) | 839 (2.5%) | 0.0% (-0.2%, 0.3%) |
|---|---|---|---|---|---|---|
| Anti-arrhythmics; n (%) Statins; n (%) | 1,631 (2.5%)<br>54,445 (83.1%) | 3,413 (2.3%)<br>116,370 (79.4%) | 3.7% (3.3%, 4.1%) | 851 (2.5%)<br>28,349 (83.4%) | 28,402 (83.6%) | -0.2% (-0.2%, 0.3%) |
| | 8,155 (12.4%) | 19,421 (13,3%) | -0.8% (-1.1%, -0.5%) | 4.514 (13.3%) | 4,569 (13,4%) | -0.2% (-0.7%, 0.4%) |
| PCSK9 inhibitors and other lipid-lowering drugs; n (%) | | | 1.5% (1.2%, 1.8%) | , | , | |
| Antiplatelet medications; n (%) | 7,633 (11.7%) | 14,864 (10.1%) | | 3,770 (11.1%)<br>3,834 (11.3%) | 3,786 (11.1%)<br>3,780 (11.1%) | -0.0% (-0.5%, 0.4%) |
| Oral anticoagulants; n (%) | 7,403 (11.3%) | 15,122 (10.3%) | 1.0% (0.7%, 1.3%) | .,, | -, - , - , | 0.2% (-0.3%, 0.6%) |
| COPD/Asthma medications; n (%) | 22,260 (34.0%) | 53,080 (36.2%) | -2.2% (-2.7%, -1.8%) | 11,961 (35.2%) | 12,093 (35.6%) | -0.4% (-1.1%, 0.3%) |
| NSAIDS; n (%) | 20,582 (31.4%) | 49,724 (33.9%) | -2.5% (-2.9%, -2.1%) | 11,262 (33.1%) | 11,367 (33.5%) | -0.3% (-1.0%, 0.4%) |
| Oral corticosteroids; n (%) | 13,316 (20.3%) | 37,969 (25.9%) | -5.6% (-6.0%, -5.2%) | 7,437 (21.9%) | 7,426 (21.9%) | 0.0% (-0.6%, 0.7%) |
| Osteoporosis agents (incl. bisphosphonates); n (%) | 2,736 (4.2%) | 3,717 (2.5%) | 1.6% (1.5%, 1.8%) | 1,209 (3.6%) | 1,197 (3.5%) | 0.0% (-0.2%, 0.3%) |
| Opioids; n (%) | 21,041 (32.1%) | 47,067 (32.1%) | 0.0% (-0.4%, 0.4%) | 10,780 (31.7%) | 10,896 (32.1%) | -0.3% (-1.0%, 0.4%) |
| Anti-depressants; n (%) | 21,685 (33.1%) | 59,566 (40.6%) | -7.5% (-8.0%, -7.1%) | 12,325 (36.3%) | 12,425 (36.6%) | -0.3% (-1.0%, 0.4%) |
| Antipsychotics; n (%) | 3,011 (4.6%) | 7,152 (4.9%) | -0.3% (-0.5%, -0.1%) | 1,618 (4.8%) | 1,683 (5.0%) | -0.2% (-0.5%, 0.1%) |
| Anxiolytics / hypnotics, benzos; n (%) | 12,831 (19.6%) | 32,904 (22.5%) | -2.9% (-3.2%, -2.5%) | 6,947 (20.4%) | 6,945 (20.4%) | 0.0% (-0.6%, 0.6%) |
| Dementia medications; n (%) | 2,314 (3.5%) | 1,819 (1.2%) | 2.3% (2.1%, 2.4%) | 828 (2.4%) | 854 (2.5%) | -0.1% (-0.3%, 0.2%) |
| Urinary tract infections antibiotics; n (%) | 30,037 (45.9%) | 68,561 (46.8%) | -0.9% (-1.4%, -0.5%) | 15,553 (45.8%) | 15,597 (45.9%) | -0.1% (-0.9%, 0.6%) |
| Laxatives; n (%) | 2,582 (3.9%) | 5,244 (3.6%) | 0.4% (0.2%, 0.5%) | 1,224 (3.6%) | 1,203 (3.5%) | 0.1% (-0.2%, 0.3%) |
| Number of distinct medications | | | | | | |
| mean (sd) | 14.62 (6.77) | 14.67 (7.03) | -0.06 (-0.12, 0.01) | 14.81 (6.91) | 14.93 (6.83) | -0.12 (-0.23, -0.02) |
| median [IQR] | 14.00 [10.00, 18.00] | 14.00 [10.00, 19.00] | - (-, -) | 14.00 [10.00, 19.00] | 14.00 [10.00, 19.00] | - (-, -) |
| min, max | 1.00, 69.00 | 1.00, 72.00 | - (-, -) | 1.00, 69.00 | 1.00, 65.00 | - (-, -) |
| Number of office visits | | | | | | |
| mean (sd) | 9.46 (6.88) | 9.79 (7.09) | -0.33 (-0.40, -0.27) | 9.61 (7.04) | 9.70 (6.82) | -0.09 (-0.20, 0.01) |
| median [IQR] | 8.00 [5.00, 13.00] | 8.00 [5.00, 13.00] | - (-, -) | 8.00 [5.00, 13.00] | 8.00 [5.00, 13.00] | - (-, -) |
| min, max | 0.00, 123.00 | 0.00, 115.00 | - (-, -) | 0.00, 93.00 | 0.00, 94.00 | - (-, -) |
| Number of endocrinologist visits | | | 17.7 | , | | 17.7 |
| mean (sd) | 0.32 (1.31) | 0.48 (1.44) | -0.16 (-0.17, -0.15) | 0.37 (1.50) | 0.39 (1.15) | -0.02 (-0.04, -0.00) |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - () | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) |
| min. max | 0.00, 65.00 | 0.00, 53.00 | - (-, -) | 0.00, 65.00 | 0.00, 23.00 | - (-, -) |
| Number of cardiologist visits | 0.00, 03.00 | 0.00, 55.00 | - (-, -) | 0.00, 03.00 | 0.00, 23.00 | - (-, -) |
| mean (sd) | 1.89 (3.93) | 1.59 (3.58) | 0.29 (0.26, 0.33) | 1.75 (3.82) | 1.76 (3.84) | -0.00 (-0.06, 0.05) |
| | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | - (-, -) | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | - (-, -) |
| median [IQR] | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | |
| min, max | 0.00, 117.00 | 0.00, 160.00 | - (-, -) | 0.00, 83.00 | 0.00, 105.00 | - (-, -) |
| Number of internal/family medicine visits | 0.00(0.00) | 7.21 (0.20) | 150 (1.47.105) | 0.21 (0.20) | 0.26 (0.60) | 0.00 ( 0.20 0.00) |
| mean (sd) | 8.86 (9.69) | 7.31 (8.36) | 1.56 (1.47, 1.65) | 8.31 (9.39) | 8.36 (9.68) | -0.06 (-0.20, 0.08) |
| median [IQR] | 6.00 [3.00, 11.00] | 5.00 [3.00, 9.00] | - (-, -) | 6.00 [3.00, 10.00] | 6.00 [3.00, 10.00] | - (-, -) |
| min, max | 0.00, 244.00 | 0.00, 233.00 | - (-, -) | 0.00, 244.00 | 0.00, 219.00 | - (-, -) |
| Number of electrocardiograms (ECG/EKG) | | | | | | |
| mean (sd) | 1.12 (1.88) | 0.95 (1.66) | 0.17 (0.16, 0.19) | 1.05 (1.83) | 1.05 (1.79) | -0.00 (-0.03, 0.02) |
| median [IQR] | 1.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | - (-, -) | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | - (-, -) |
| min, max | 0.00, 42.00 | 0.00, 48.00 | - (-, -) | 0.00, 42.00 | 0.00, 48.00 | - (-, -) |
| Number of echocardiograms | | | | | | |
| mean (sd) | 0.32 (0.67) | 0.28 (0.64) | 0.04 (0.03, 0.05) | 0.30 (0.66) | 0.30 (0.65) | 0.00 (-0.01, 0.01) |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) |
| min, max | 0.00, 12.00 | 0.00, 24.00 | - (-, -) | 0.00, 12.00 | 0.00, 9.00 | - (-, -) |
| Out-of-pocket medication cost | | | | | | |
| mean (sd) | 528.48 (675.73) | 589.31 (766.63) | -60.83 (-67.33, -54.34) | 549.80 (736.21) | 556.67 (619.95) | -6.87 (-17.10, 3.37) |
| median [IQR] | 300.20 [118.88, 700.12] | 349.61 [140.87, 783.39] | - (-, -) | 295.08 [116.23, 730.45] | 346.20 [143.12, 756.61] | - (-, -) |
| min, max | 0.00, 27,404.93 | 0.00, 51,242.99 | - (-, -) | 0.00, 27,404.93 | 0.00, 14,359.16 | - (-, -) |
| Unique brand medicines | | | | | | |
| mean (sd) | 14.88 (7.01) | 14.97 (7.27) | -0.08 (-0.15, -0.02) | 15.09 (7.16) | 15.22 (7.07) | -0.13 (-0.23, -0.02) |
| median [IQR] | 14.00 [10.00, 19.00] | 14.00 [10.00, 19.00] | - (-, -) | 14.00 [10.00, 19.00] | 14.00 [10.00, 19.00] | - (-, -) |
| min, max | 1.00, 74.00 | 1.00, 84.00 | - (-, -) | 1.00, 74.00 | 1.00, 69.00 | - (-, -) |
| Unique generic medicines | | | 377 | | | (1) |
| mean (sd) | 14.62 (6.77) | 14.67 (7.03) | -0.06 (-0.12, 0.01) | 14.81 (6.91) | 14.93 (6.83) | -0.12 (-0.23, -0.02) |
| median [IQR] | 14.00 [10.00, 18.00] | 14.00 [10.00, 19.00] | - (-, -) | 14.00 [10.00, 19.00] | 14.00 [10.00, 19.00] | - (-, -) |
| min. max | 1.00, 69.00 | 1.00, 72.00 | - (-, -)<br>- (-, -) | 1.00, 69.00 | 1.00, 65.00 | - (-, -) |
| Colonoscopy Sigmoidoscopy; n (%) | 6,142 (9.4%) | 15,505 (10.6%) | -1.2% (-1.5%, -0.9%) | 3,348 (9.9%) | 3,330 (9.8%) | 0.1% (-0.4%, 0.5%) |
| | 6,142 (9.4%)<br>25,667 (39.2%) | | -1.2% (-1.5%, -0.9%)<br>5.6% (5.1%, 6.0%) | 12,484 (36.7%) | | -0.1% (-0.4%, 0.5%) |
| Flu Pneumococcal vaccine; n (%) | | 49,218 (33.6%) | | | 12,513 (36.8%) | |
| Pap smear, n (%) | 2,812 (4.3%) | 11,052 (7.5%) | -3.2% (-3.5%, -3.0%) | 1,649 (4.9%) | 1,643 (4.8%) | 0.0% (-0.3%, 0.3%) |
| PSA test; n (%) | 14,180 (21.6%) | 31,754 (21.7%) | -0.0% (-0.4%, 0.4%) | 7,400 (21.8%) | 7,375 (21.7%) | 0.1% (-0.5%, 0.7%) |
| Fecal occult blood test; n (%) | 5,592 (8.5%) | 6,401 (4.4%) | 4.2% (3.9%, 4.4%) | 2,186 (6.4%) | 2,191 (6.4%) | -0.0% (-0.4%, 0.4%) |
| Bone mineral density tests; n (%) | 5,684 (8.7%) | 10,824 (7.4%) | 1.3% (1.0%, 1.5%) | 2,898 (8.5%) | 2,864 (8.4%) | 0.1% (-0.3%, 0.5%) |
| Mammograms; n (%) | 15,397 (23.5%) | 39,540 (27.0%) | -3.5% (-3.9%, -3.1%) | 8,582 (25.3%) | 8,558 (25.2%) | 0.1% (-0.6%, 0.7%) |
| Telemedicine; n (%) | 10,567 (16.1%) | 37,986 (25.9%) | -9.8% (-10.2%, -9.4%) | 7,496 (22.1%) | 7,599 (22.4%) | -0.3% (-0.9%, 0.3%) |
| HbA1c tests | | | | | <u> </u> | |

| mean (sd) | 2.42 (1.34) | 2.34 (1.33) | 0.08 (0.06, 0.09) | 2.41 (1.34) | 2.43 (1.34) | -0.02 (-0.04, 0.00) |
|---|---|---|---|---|---|---|
| median [IQR] | 2.00 [2.00, 3.00] | 2.00 [1.00, 3.00] | - (-, -) | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | - (-, -) |
| min, max | 0.00, 50.00 | 0.00, 75.00 | - (-, -) | 0.00, 50.00 | 0.00, 34.00 | - (-, -) |
| Lipid panels | | | | | | |
| mean (sd) | 1.70 (1.20) | 1.64 (1.18) | 0.06 (0.05, 0.07) | 1.68 (1.18) | 1.67 (1.16) | 0.01 (-0.01, 0.03) |
| median [IQR] | 2.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | - (-, -) | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | - (-, -) |
| min, max | 0.00, 27.00 | 0.00, 75.00 | - (-, -) | 0.00, 27.00 | 0.00, 31.00 | - (-, -) |
| Creatinine tests | | | | | | |
| mean (sd) | 3.21 (3.19) | 2.87 (2.90) | 0.35 (0.32, 0.37) | 3.14 (3.33) | 3.15 (3.27) | -0.01 (-0.06, 0.04) |
| median [IQR] | 3.00 [2.00, 4.00] | 2.00 [1.00, 4.00] | - (-, -) | 3.00 [1.00, 4.00] | 3.00 [1.00, 4.00] | - (-, -) |
| min, max | 0.00, 366.00 | 0.00, 118.00 | - (-, -) | 0.00, 366.00 | 0.00, 118.00 | - (-, -) |
| Natriuretic peptide tests | | | | | | |
| mean (sd) | 0.19 (1.59) | 0.18 (0.79) | 0.01 (-0.01, 0.02) | 0.19 (2.10) | 0.19 (0.67) | 0.01 (-0.02, 0.03) |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) |
| min, max | 0.00, 366.00 | 0.00, 77.00 | - (-, -) | 0.00, 366.00 | 0.00, 18.00 | - (-, -) |
| Urine tests | | | | | | |
| mean (sd) | 1.25 (2.28) | 1.04 (1.64) | 0.21 (0.19, 0.23) | 1.17 (2.62) | 1.17 (1.80) | 0.00 (-0.03, 0.04) |
| median [IQR] | 1.00 [0.00, 2.00] | 0.00 [0.00, 1.00] | - (-, -) | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | - (-, -) |
| min, max | 0.00, 366.00 | 0.00, 73.00 | - (-, -) | 0.00, 366.00 | 0.00, 73.00 | - (-, -) |
| Combined comorbidity score | | | | | | |
| mean (sd) | 2.62 (2.77) | 1.96 (2.38) | 0.66 (0.63, 0.68) | 2.35 (2.58) | 2.37 (2.62) | -0.02 (-0.06, 0.02) |
| median [IQR] | 2.00 [1.00, 4.00] | 1.00 [0.00, 3.00] | - (-, -) | 2.00 [0.00, 4.00] | 2.00 [0.00, 4.00] | - (-, -) |
| min, max | -2.00, 17.00 | -2.00, 16.00 | - (-, -) | -2.00, 16.00 | -2.00, 16.00 | - (-, -) |
| Frailty Score | | | | | | |
| mean (sd) | 0.18 (0.06) | 0.17 (0.06) | 0.01 (0.01, 0.01) | 0.17 (0.06) | 0.17 (0.06) | -0.00 (-0.00, 0.00) |
| median [IQR] | 0.17 [0.13, 0.21] | 0.16 [0.13, 0.19] | - (-, -) | 0.16 [0.13, 0.20] | 0.16 [0.13, 0.20] | - (-, -) |
| min, max | 0.03, 0.67 | 0.03, 0.62 | - (-, -) | 0.03, 0.62 | 0.04, 0.62 | - (-, -) |
| Number of Hospitalizations | | | | | | |
| mean (sd) | 0.33 (0.96) | 0.20 (0.65) | 0.14 (0.13, 0.15) | 0.27 (0.84) | 0.27 (0.85) | -0.00 (-0.01, 0.01) |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) |
| min, max | 0.00, 29.00 | 0.00, 26.00 | - (-, -) | 0.00, 27.00 | 0.00, 26.00 | - (-, -) |
| Any hospitalization within prior 91 days; n (%) | 5,714 (8.7%) | 6,298 (4.3%) | 4.4% (4.2%, 4.7%) | 2,192 (6.5%) | 2,238 (6.6%) | -0.1% (-0.5%, 0.2%) |
| Any hospitalization within prior 92-365 days; n (%) | 8,358 (12.8%) | 14,569 (9.9%) | 2.8% (2.5%, 3.1%) | 3,889 (11.4%) | 3,899 (11.5%) | -0.0% (-0.5%, 0.5%) |
| Number of hospitalizations (0, 1, 2 or more) | | | | | | |
| < 1; n (%) | 53,635 (81.9%) | 127,957 (87.3%) | -5.4% (-5.8%, -5.1%) | 28,752 (84.6%) | 28,746 (84.6%) | 0.0% (-0.5%, 0.6%) |
| 1 - <2; n (%) | 7,022 (10.7%) | 12,994 (8.9%) | 1.9% (1.6%, 2.1%) | 3,294 (9.7%) | 3,279 (9.7%) | 0.0% (-0.4%, 0.5%) |
| >= 2; n (%) | 4,852 (7.4%) | 5,589 (3.8%) | 3.6% (3.4%, 3.8%) | 1,927 (5.7%) | 1,948 (5.7%) | -0.1% (-0.4%, 0.3%) |
| Heart failure hospitalization; n (%) | 3,416 (5.2%) | 5,056 (3.5%) | 1.8% (1.6%, 2.0%) | 1,491 (4.4%) | 1,448 (4.3%) | 0.1% (-0.2%, 0.4%) |
| ED visit; n (%) | 24,198 (36.9%) | 41,255 (28.2%) | 8.8% (8.3%, 9.2%) | 11,600 (34.1%) | 11,610 (34.2%) | -0.0% (-0.7%, 0.7%) |
| Acute MI; n (%) | 877 (1.3%) | 1,628 (1.1%) | 0.2% (0.1%, 0.3%) | 406 (1.2%) | 419 (1.2%) | -0.0% (-0.2%, 0.1%) |
| Old MI; n (%) | 3,762 (5.7%) | 6,389 (4.4%) | 1.4% (1.2%, 1.6%) | 1,756 (5.2%) | 1,729 (5.1%) | 0.1% (-0.3%, 0.4%) |
| Heart failure; n (%) | 10,742 (16.4%) | 19,955 (13.6%) | 2.8% (2.4%, 3.1%) | 5,219 (15.4%) | 5,254 (15.5%) | -0.1% (-0.6%, 0.4%) |
| Acute heart failure; n (%) | 2,954 (4.5%) | 4,816 (3.3%) | 1.2% (1.0%, 1.4%) | 1,334 (3.9%) | 1,319 (3.9%) | 0.0% (-0.3%, 0.3%) |
| Microalbuminuria or proteinuria; n (%) | 4,267 (6.5%) | 9,587 (6.5%) | -0.0% (-0.3%, 0.2%) | 2,173 (6.4%) | 2,198 (6.5%) | -0.1% (-0.4%, 0.3%) |
| Ratio of brand to generic medications | | | | | | |
| mean (sd) | 1.02 (0.04) | 1.02 (0.04) | -0.00 (-0.00, -0.00) | 1.02 (0.04) | 1.02 (0.04) | -0.00 (-0.00, 0.00) |
| median [IQR] | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | - (-, -) | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | - (-, -) |
| min, max | 0.80, 2.00 | 0.80, 1.83 | - (-, -) | 0.80, 2.00 | 0.85, 1.42 | - (-, -) |
| <b>-</b> | | | | | | |

Appendix 7. Balance Assessment - Table 1

| MARKETSCAN | | | | | | |
|---|---|---|---|---|---|---|
| Variable | Reference: Sitagliptin | Exposure: Semaglutide injection | Difference | Reference: Sitagliptin | Exposure: Semaglutide injection | Difference |
| Number of patients | 62,457 | 100,869 | - (-, -) | 33,189 | 33,189 | - (-, -) |
| Year of Cohort Entry Date | 02,437 | 100,003 | ( , ) | 33,103 | 33,103 | ( , ) |
| 2018: n (%) | 16.154 (25.9%) | 2.333 (2.3%) | 23.6% (23.2%, 23.9%) | 2.254 (6.8%) | 2.274 (6.9%) | -0.1% (-0.4%, 0.3%) |
| 2019; n (%) | 14,495 (23.2%) | 8,407 (8.3%) | 14.9% (14.5%, 15.2%) | 6,554 (19.7%) | 6,664 (20.1%) | -0.3% (-0.9%, 0.3%) |
| 2020; n (%) | 11,269 (18.0%) | | 8.2% (7.9%, 8.6%) | 6,697 (20.2%) | 6,730 (20.3%) | -0.1% (-0.7%, 0.5%) |
| 2021; n (%) | 9,490 (15.2%) | 15,532 (15.4%) | -0.2% (-0.6%, 0.2%) | 7,370 (22.2%) | 7,371 (22.2%) | -0.0% (-0.6%, 0.6%) |
| 2022; n(%) | 6,420 (10,3%) | 22,846 (22.6%) | -12.4% (-12.7%, -12.0%) | 5,840 (17.6%) | 5,780 (17,4%) | 0.2% (-0.4%, 0.8%) |
| 2023; n (%) | 4.629 (7.4%) | 41.836 (41.5%) | -34.1% (-34.4%, -33.7%) | 4,474 (13.5%) | 4,370 (13.2%) | 0.3% (-0.2%, 0.8%) |
| Age | 1,020 (7.170) | 12,000 (12070) | 0 11270 ( 0 11 170) ( 00.770) | 1,171 (25.676) | 1,070 (10.1270) | 0.070 ( 0.270, 0.070) |
| mean (sd) | 57.85 (11.72) | 53.66 (9.98) | 4.19 (4.08, 4.30) | 55.50 (11.21) | 55.51 (9.68) | -0.00 (-0.16, 0.15) |
| median [IQR] | 58.00 [50.00, 64.00] | 54.00 [47.00, 60.00] | - (-, -) | 56.00 [48.00, 62.00] | 56.00 [49.00, 61.00] | - (-, -) |
| min, max | 18.00, 99.00 | 18.00, 95.00 | - (-, -) | 18.00, 97.00 | 18.00, 95.00 | - (-, -) |
| Gender (male); n (%) | 32,670 (52.3%) | 45,429 (45.0%) | 7.3% (6.8%, 7.8%) | 16,431 (49.5%) | 16,431 (49.5%) | 0.0% (-0.8%, 0.8%) |
| Region / State | , | | | ., | | |
| Northeast; n (%) | 10,524 (16.8%) | 11,928 (11.8%) | 5.0% (4.7%, 5.4%) | 4,897 (14.8%) | 4,827 (14.5%) | 0.2% (-0.3%, 0.8%) |
| Widwest / North central; n (%) | 16,026 (25.7%) | 20,650 (20.5%) | 5.2% (4.8%, 5.6%) | 7,415 (22.3%) | 7,344 (22.1%) | 0.2% (-0.4%, 0.8%) |
| South; n (%) | 31,366 (50.2%) | 59,129 (58.6%) | -8.4% (-8.9%, -7.9%) | 18,355 (55.3%) | 18,418 (55.5%) | -0.2% (-0.9%, 0.6%) |
| West; n (%) | 4,434 (7.1%) | 9,066 (9.0%) | -1.9% (-2.2%, -1.6%) | 2,479 (7.5%) | 2,559 (7.7%) | -0.2% (-0.6%, 0.2%) |
| Missing; n (%) | 107 (0.2%) | 96 (0.1%) | 0.1% (0.0%, 0.1%) | 43 (0.1%) | 41 (0.1%) | 0.0% (-0.1%, 0.1%) |
| Smoking / Tobacco use; n (%) | 6,486 (10.4%) | | 0.6% (0.3%, 0.9%) | 3,336 (10.1%) | 3,338 (10.1%) | -0.0% (-0.5%, 0.5%) |
| Weight | -, (, | -,,, | | -, (, | -,, | |
| Underweight; n (%) | 37 (0.1%) | 37 (0.0%) | 0.0% (-0.0%, 0.0%) | 14 (0.0%) | 20 (0.1%) | -0.0% (-0.1%, 0.0%) |
| Normal weight; n (%) | 516 (0.8%) | 199 (0.2%) | 0.6% (0.6%, 0.7%) | 143 (0.4%) | 148 (0.4%) | -0.0% (-0.1%, 0.1%) |
| Overweight; n (%) | 11,877 (19.0%) | | 10.6% (10.3%, 11.0%) | 4,432 (13.4%) | 4,509 (13.6%) | -0.2% (-0.8%, 0.3%) |
| Class 1 Obesity; n (%) | 8,213 (13.1%) | 8,446 (8.4%) | 4.8% (4.5%, 5.1%) | 3,714 (11.2%) | 3,747 (11.3%) | -0.1% (-0.6%, 0.4%) |
| Class 2 Obesity; n (%) | 4,739 (7.6%) | 7,022 (7.0%) | 0.6% (0.4%, 0.9%) | 2,577 (7.8%) | 2,577 (7.8%) | 0.0% (-0.4%, 0.4%) |
| Class 3 Obesity; n (%) | 15,207 (24.3%) | 30,309 (30.0%) | -5.7% (-6.1%, -5.3%) | 9,802 (29.5%) | 9,875 (29.8%) | -0.2% (-0.9%, 0.5%) |
| Unspecified Obesity; n (%) | 21,868 (35.0%) | 46,402 (46.0%) | -11.0% (-11.5%, -10.5%) | 12,507 (37.7%) | 12,313 (37.1%) | 0.6% (-0.2%, 1.3%) |
| Diabetic retinopathy; n (%) | 3,779 (6.1%) | 5,532 (5.5%) | 0.6% (0.3%, 0.8%) | 1,906 (5.7%) | 1,970 (5.9%) | -0.2% (-0.6%, 0.2%) |
| Diabetic neuropathy; n (%) | 10,029 (16.1%) | 14,342 (14.2%) | 1.8% (1.5%, 2.2%) | 5,062 (15.3%) | 5,082 (15.3%) | -0.1% (-0.6%, 0.5%) |
| Diabetic nephropathy; n (%) | 7,446 (11.9%) | 10,355 (10.3%) | 1.7% (1.3%, 2.0%) | 3,623 (10.9%) | 3,791 (11.4%) | -0.5% (-1.0%, -0.0%) |
| Diabetes with other opthalmic complications; n (%) | 929 (1.5%) | 1,336 (1.3%) | 0.2% (0.0%, 0.3%) | 484 (1.5%) | 488 (1.5%) | -0.0% (-0.2%, 0.2%) |
| Diabetes with peripheral circulatory disorders; n (%) | 3,938 (6.3%) | 6,575 (6.5%) | -0.2% (-0.5%, 0.0%) | 2,023 (6.1%) | 2,062 (6.2%) | -0.1% (-0.5%, 0.3%) |
| Diabetic foot; n (%) | 1,033 (1.7%) | 1,519 (1.5%) | 0.1% (0.0%, 0.3%) | 511 (1.5%) | 497 (1.5%) | 0.0% (-0.1%, 0.2%) |
| Erectile dysfunction; n (%) | 2,436 (3.9%) | 3,749 (3.7%) | 0.2% (-0.0%, 0.4%) | 1,300 (3.9%) | 1,337 (4.0%) | -0.1% (-0.4%, 0.2%) |
| Hypoglycemia; n (%) | 7,914 (12.7%) | 16,135 (16.0%) | -3.3% (-3.7%, -3.0%) | 4,631 (14.0%) | 4,648 (14.0%) | -0.1% (-0.6%, 0.5%) |
| Hyperglycemia/DKA/HONK; n (%) | 30,989 (49.6%) | 50,576 (50.1%) | -0.5% (-1.0%, -0.0%) | 17,026 (51.3%) | 17,227 (51.9%) | -0.6% (-1.4%, 0.2%) |
| Skin infections; n (%) | 5,552 (8.9%) | 8,922 (8.8%) | 0.0% (-0.2%, 0.3%) | 2,954 (8.9%) | 2,990 (9.0%) | -0.1% (-0.5%, 0.3%) |
| Stable angina; n (%) | 1,440 (2.3%) | 2,179 (2.2%) | 0.1% (-0.0%, 0.3%) | 737 (2.2%) | 757 (2.3%) | -0.1% (-0.3%, 0.2%) |
| Unstable angina; n (%) | 1,143 (1.8%) | 1,554 (1.5%) | 0.3% (0.2%, 0.4%) | 538 (1.6%) | 545 (1.6%) | -0.0% (-0.2%, 0.2%) |
| Hypertension; n (%) | 51,108 (81.8%) | 80,690 (80.0%) | 1.8% (1.4%, 2.2%) | 26,797 (80.7%) | 26,784 (80.7%) | 0.0% (-0.6%, 0.6%) |
| Hypotension; n (%) | 1,071 (1.7%) | 1,289 (1.3%) | 0.4% (0.3%, 0.6%) | 482 (1.5%) | 472 (1.4%) | 0.0% (-0.2%, 0.2%) |
| Hyperlipidemia; n (%) | 49,887 (79.9%) | 78,385 (77.7%) | 2.2% (1.8%, 2.6%) | 26,306 (79.3%) | 26,364 (79.4%) | -0.2% (-0.8%, 0.4%) |
| Atrial fibrillation; n (%) | 3,601 (5.8%) | 4,460 (4.4%) | 1.3% (1.1%, 1.6%) | 1,568 (4.7%) | 1,558 (4.7%) | 0.0% (-0.3%, 0.4%) |
| Cardiac conduction disorder; n (%) | 1,831 (2.9%) | | 0.4% (0.2%, 0.6%) | 830 (2.5%) | 846 (2.5%) | -0.0% (-0.3%, 0.2%) |
| Previous cardiac procedure (CABG, PTCA, Stent); n (%) | 821 (1.3%) | 1,238 (1.2%) | 0.1% (-0.0%, 0.2%) | 421 (1.3%) | 446 (1.3%) | -0.1% (-0.3%, 0.1%) |
| Ischemic stroke; n (%) | 716 (1.1%) | 709 (0.7%) | 0.4% (0.3%, 0.5%) | 268 (0.8%) | 276 (0.8%) | -0.0% (-0.2%, 0.1%) |
| PVD diagnosis or surgery; n (%) | 3,073 (4.9%) | | 1.6% (1.4%, 1.9%) | 1,268 (3.8%) | 1,299 (3.9%) | -0.1% (-0.4%, 0.2%) |
| Other cardiac dysrhythmia; n (%) | 8,337 (13.3%) | 13,698 (13.6%) | -0.2% (-0.6%, 0.1%) | 4,225 (12.7%) | 4,214 (12.7%) | 0.0% (-0.5%, 0.5%) |
| Cardiomyopathy; n (%) | 1,851 (3.0%) | | 0.4% (0.2%, 0.5%) | 841 (2.5%) | 874 (2.6%) | -0.1% (-0.3%, 0.1%) |
| Valve disorders; n (%) | 3,978 (6.4%) | 5,470 (5.4%) | 0.9% (0.7%, 1.2%) | 1,840 (5.5%) | 1,843 (5.6%) | -0.0% (-0.4%, 0.3%) |
| Valve replacement; n (%) | 377 (0.6%) | 433 (0.4%) | 0.2% (0.1%, 0.2%) | 142 (0.4%) | 150 (0.5%) | -0.0% (-0.1%, 0.1%) |
| TIA; n (%) | 858 (1.4%) | | 0.4% (0.2%, 0.5%) | 372 (1.1%) | 364 (1.1%) | 0.0% (-0.1%, 0.2%) |
| Edema; n (%) | 4,489 (7.2%) | 7,624 (7.6%) | -0.4% (-0.6%, -0.1%) | 2,310 (7.0%) | 2,314 (7.0%) | -0.0% (-0.4%, 0.4%) |
| Venous thromboembolism / Pulmonary embolism; n (%) | 1,419 (2.3%) | | 0.1% (-0.1%, 0.2%) | 709 (2.1%) | 685 (2.1%) | 0.1% (-0.1%, 0.3%) |
| Pulmonary hypertension; n (%) | 784 (1.3%) | 1,064 (1.1%) | 0.2% (0.1%, 0.3%) | 357 (1.1%) | 344 (1.0%) | 0.0% (-0.1%, 0.2%) |
| Implantable cardioverter defibrillator; n (%) | 111 (0.2%) | 164 (0.2%) | 0.0% (-0.0%, 0.1%) | 52 (0.2%) | 56 (0.2%) | -0.0% (-0.1%, 0.1%) |
| Hyperkalemia; n (%) | 1,020 (1.6%) | | 0.4% (0.3%, 0.5%) | 455 (1.4%) | 486 (1.5%) | -0.1% (-0.3%, 0.1%) |
| Coronary atherosclerosis; n (%) | 8,059 (12.9%) | 10,879 (10.8%) | 2.1% (1.8%, 2.4%) | 3,692 (11.1%) | 3,803 (11.5%) | -0.3% (-0.8%, 0.2%) |
| Cerebrovascular procedure; n (%) | 52 (0.1%) | 54 (0.1%) | 0.0% (0.0%, 0.1%) | 15 (0.0%) | 23 (0.1%) | -0.0% (-0.1%, 0.0%) |
| Insertion of pacemakers / removal of cardiac lead; n (%) | 59 (0.1%) | 43 (0.0%) | 0.1% (0.0%, 0.1%) | 16 (0.0%) | 19 (0.1%) | -0.0% (-0.0%, 0.0%) |
| CKD stage 1-2; n (%) | 1,356 (2.2%) | 1,896 (1.9%) | 0.3% (0.1%, 0.4%) | 648 (2.0%) | 660 (2.0%) | -0.0% (-0.3%, 0.2%) |

| Important Colon Print | CKD stage 3-4; n (%) | 3.936 (6.3%) | 4.484 (4.4%) | 1.9% (1.6%, 2.1%) | 1.697 (5.1%) | 1.721 (5.2%) | -0.1% (-0.4%, 0.3%) |
|---|---|---|---|---|---|---|---|
| Anna France (1997) Anna Fr | | .,, | | | , | | |
| Importance settlementary of 19 | | | | | | | |
| Comp petiting from (19) | | | | | | | |
| Contact Internation | | | | | | | |
| Content | | | | | | | |
| CORPORTING 1,861,6509 | | | | | | | |
| Semonth | | | | | | | |
| Distriction (Control Control | | | | | | | |
| Settle | | | | | | | |
| Pasentine Pase | | | | | | | |
| Lord States (Ling Ling State Ling Stat | | | | | | | |
| MASH MASH Direct Mash Ma | | | | | | / - / - / | |
| Parkers (PS) | | | | | | | |
| Dissemblering (Pil) | | | | | | | |
| Discontinist (CP) | | | | | | | |
| Dependent (PN) 1,259 (1,27%) 1,258 (1,17%) 1,258 (1,17%) 3.91 (1,27%) | | | | | | | |
| Demonster (PN) | | | | | | | |
| Dilation or psychostics (Ps) 038 (0594) 038 (0594) 038 (0594) 038 (0594) 039 (0594) | | | | | | | |
| Aceter Phi Super developer Phi Super developer Aceter | | | | | | | |
| Stage discretes (1%) | | | | | | | |
| American (%) | | | | | | | |
| Influences (16) | | | | | | | -0.1% (-0.7%, 0.6%) |
| COVID N | | | | | | | |
| Hypertyroidem: and other flyroid gland disorders: (19) 11945 (1919) 2.154 (2.24%) 2.2% (2.6%, 1.8%) 6.504 (19.9%) 6.554 (19.9%) 0.1% (0.5%, 0.7%) | | | | | | | |
| Injustry ordering (1%) | | | | | | | |
| Neghrotic syndromen (16) | | | 7 | | | | |
| Unitary incontrasence in (%) | | | | | | | |
| Billary diseases (11%) 235 (0.4%) 236 (0.2%) 134 (0.1%) 0.1% (0.1%, 0.2%) 50 (0.2%) 50 (0.2%) -0.0% (-0.1%, 0.1%) | | | | | | | |
| Parcentalistic n Phi | | | | | | | |
| Sower destruction in (19) 99 (0.2%) 114 (0.1%) 0.0% (0.0%, 0.1%) 35 (0.1%) 38 (0.1%) -0.0% (0.1%, 0.1%) 36 (0.1%) 36 (0.1%) -0.0% (0.1%, 0.1%) 38 (0.1%) -0.0% (0.1%, 0.1%) 38 (0.1%) -0.0% (0.1%, 0.1%) 38 (0.1%) -0.0% (0.1%, 0.1%) | | | | | | | |
| Castrogramis: n (%) | | | | | | | |
| Number of artifidabetic charge on CED | | | | | | | |
| Imman | | 330 (6.376) | 457 (0.570) | 0.070 ( 0.070, 0.170) | 10+ (0.070) | 200 (0.070) | 0.070 ( 0.270, 0.170) |
| Immedian (IQRI | | 2 21 (0.82) | 2.06 (0.91) | 0.14 (0.13, 0.15) | 219 (0.85) | 2 20 (0 90) | -0.02(-0.03 -0.00) |
| Imple Impl | | | | | | | |
| Concomitant use or initiation of Metromire, 1(%) | | | | | | | |
| Concomitant use or initiation of Issulins; n (%) | | | | | | | |
| Concomitant use or initiation of Sulf royluresis; n (%) 15.070 (24.1%) 13.292 (13.2%) 1.0% (10.6%; 11.3%) 6.445 (19.4%) 6.481 (19.5%) 0.1% (-0.7%) 0.5 (-0.5%) 0.5 (-0 | | | | | | | |
| Concomitant use or initiation of SQLT-2t; n (%) 5.0% (5.4%, 4.6%) 5.572 (16.8%) 5.510 (17.5%) 0.7% (1.3%, 0.1%) 0. | | ., | | | | , | |
| Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metromirin, n (%) 47,787 (76.5%) 72,578 (72.0%) 4,786 (76.5%) 72,578 (72.0%) 4,6% (4.1%, 5.0%) 25,388 (76.5%) 25,16 (76.6%) 0.1% (-0.7%, 0.6 Past use of Insulins; n (%) 8,387 (13.4%) 19,264 (12.5%) 19,10 (-9.4%, 8.7%) 19,234 (19.1%) 10,20 (12.6%) 10,400 (12.6%) 10,400 (13.6%) 10,4 | | | | | | | |
| Past use of Metformitrin (%) Past use of Insulins; n (%) B, 337 (13.4%) 22.691 (22.5%) 9.1% (9.4%, -8.7%) 5.913 (17.8%) 6.184 (18.6%) 9.254 (19.1%) 19.775 (31.7%) 19.224 (19.1%) 12.694 (12.2%, 13.0%) 8.806 (25.5%) 8.834 (26.6%) 9.184 (16.6%) 9.284 (19.1%) 9.284 (19.1%) 1.402 (18.3%) 1.402 (18.3%) 1.402 (18.3%) 1.403 (18.3%) 1.403 (18.3%) 1.403 (18.3%) 1.403 (18.3%) 1.403 (18.3%) 1.53% (5.7%, 4.9%) 1.7508 (22.6%) 1.751 (23.4%) 9.284 (6.9%) 1.761 (23.4%) 9.284 (6.9%) 1.761 (23.4%) 9.284 (6.9%) 1.761 (23.4%) 9.284 (6.9%) 1.761 (23.4%) 9.284 (6.9%) 1.761 (23.4%) 9.284 (6.9%) 9.284 (6.9%) 9.284 (6.9%) 9.285 (6.9%) 9.285 (6.9%) 9.285 (6.9%) 9.285 (6.9%) 9.286 (6.9%) 9.287 (6.9%) 9.288 (7.9%) | | | | | | | -0.1% (-0.4%, 0.2%) |
| Past use of Insulins; n (%) | | | | | | | |
| Past use of Sulfonylureas; n (%) 19,775 (31.7%) 19,234 (19.1%) 12.6% (12.2%, 13.0%) 8,806 (26.5%) 8,834 (26.6%) 0.1% (0.8%, 0.6 Past use of Sol.1-2r, n (%) 11.402 (18.3%) 23,796 (23.6%) 5.5.3% (5.7%, 4.9%) 7,508 (22.6%) 7,761 (23.4%) 0.0.8% (1.4%, 0.0.8%) 0.0.8% (1.4.8%) | | | | | | | |
| Past use of SGLT-2; n (%) | | | | | | | 0.070 ( 2.170, 0.270) |
| Past use of Any other glucose-lowering drugs; n (%) | | | | 12 6% (12 2% 13 0%) | 8 806 (26 5%) | 8 834 (26 6%) | -0.1% (-0.8%, 0.6%) |
| ACE-is/ARB's; n (%) 46,356 (74.2%) 70,619 (70.0%) 4.2% (3.8%, 4.7%) 24,113 (72.7%) 24,155 (72.8%) 0.1% (-0.8%, 0.6 ARNI; n (%) 352 (0.6%) 1,029 (1.0%) -0.5% (-0.5%, 0.4%) 221 (0.7%) 225 (0.7%) -0.0% (-0.1%, 0.6 ARNI; n (%) 20,945 (33.5%) 31,879 (31.6%) 20,935 (33.5%) 31,879 (31.6%) 1,9% (1.4%, 2.4%) 1,050 (4.31.6%) 1,052 (3.1.7%) 1,054 (3.1.6%) 1,054 (3.1.6%) 1,052 (72.7%) 1,054 (3.1.6%) 1,052 (72.7%) 1,054 (3.1.6%) 1,052 (72.7%) 1,054 (3.1.6%) 1,052 (72.7%) 1,054 (3.1.6%) | | | | | | | -0.1% (-0.8%, 0.6%)<br>-0.8% (-1.4%, -0.1%) |
| ARNI; n (%) | Past use of SGLT-2i; n (%) | 11,402 (18.3%) | 23,796 (23.6%) | -5.3% (-5.7%, -4.9%) | 7,508 (22.6%) | 7,761 (23.4%) | -0.1% (-0.8%, 0.6%)<br>-0.8% (-1.4%, -0.1%)<br>-0.1% (-0.5%, 0.3%) |
| Thiazides; n (%) 20,945 (33.5%) 35,859 (35.6%) 20% (-2.5%, -1.5%) 11,443 (34.5%) 11,415 (34.4%) 0.1% (-0.6%, 0.8 Beta-blockers; n (%) 20,935 (33.5%) 31,879 (31.6%) 1.9% (1.4%, 2.4%) 10,504 (31.6%) 10,528 (31.7%) -0.1% (-0.8%, 0.8 Deta-blockers; n (%) 18,193 (29.1%) 27,539 (27.3%) 1.8% (1.4%, 2.3%) 9,267 (27.9%) 9,183 (27.7%) 0.3% (-0.4%, 0.2 Degxin / Digitoxin; n (%) 366 (0.6%) 309 (0.3%) 0.3% (0.2%, 0.3%) 137 (0.4%) 136 (0.4%) 0.0% (-0.1%, 0.1% (-0.5%, 0.1 Degxin / Digitoxin; n (%) 136 (0.4%) 0.0% (-0.5%, 0.1 Degxin / Digitoxin; n (%) 137 (0.4%) 136 (0.4%) 0.0% (-0.5%, 0.1 Degxin / Digitoxin; n (%) 137 (0.4%) 137 (0.4%) 137 (0.4%) 137 (0.4%) 136 (0.4%) 0.0% (-0.5%, 0.1 Degxin / Digitoxin; n (%) 137 (0.4%) | Past use of SGLT-2i; n (%) Past use of Any other glucose-lowering drugs; n (%) | 11,402 (18.3%)<br>4,351 (7.0%) | 23,796 (23.6%)<br>5,580 (5.5%) | -5.3% (-5.7%, -4.9%)<br>1.4% (1.2%, 1.7%) | 7,508 (22.6%)<br>2,242 (6.8%) | 7,761 (23.4%)<br>2,280 (6.9%) | -0.8% (-1.4%, -0.1%) |
| Beta-blockers; n (%) 20,935 (33.5%) 31,879 (31.6%) 1,9% (1.4%, 2.4%) 10,504 (31.6%) 10,528 (31.7%) -0.1% (-0.8%, 0.6 | Past use of SGLT-2i; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) | 11,402 (18.3%)<br>4,351 (7.0%)<br>46,356 (74.2%) | 23,796 (23.6%)<br>5,580 (5.5%)<br>70,619 (70.0%) | -5.3% (-5.7%, -4.9%)<br>1.4% (1.2%, 1.7%)<br>4.2% (3.8%, 4.7%) | 7,508 (22.6%)<br>2,242 (6.8%)<br>24,113 (72.7%) | 7,761 (23.4%)<br>2,280 (6.9%)<br>24,155 (72.8%) | -0.8% (-1.4%, -0.1%)<br>-0.1% (-0.5%, 0.3%)<br>-0.1% (-0.8%, 0.6%) |
| Calcium channel blockers; $n$ (%) 18,193 (29.1%) 27,539 (27.3%) 1.8% (1.4%, 2.3%) 9,267 (27.9%) 9,183 (27.7%) 0.3% (-0.4%, 0.5%) Digoxin / Digitoxin; $n$ (%) 366 (0.6%) 309 (0.3%) 0.3% (0.2%, 0.3%) 137 (0.4%) 136 (0.4%) 0.0% (-0.1%, 0.1%) Loop directics; $n$ (%) 6,024 (9.6%) 9,811 (9.7%) -0.1% (-0.4%, 0.2%) 3,005 (9.1%) 3,016 (9.1%) -0.0% (-0.5%, 0.2%) Other diuretics; $n$ (%) 3,731 (6.0%) 7,652 (7.6%) -1.6% (1.9%, -1.4%) 2.092 (6.3%) 2,148 (6.5%) -0.2% (-0.5%, 0.2%) Intravenous diuretics; $n$ (%) 331 (0.5%) 565 (0.6%) -0.0% (-0.1%, 0.0%) 153 (0.5%) 154 (0.5%) -0.0% (-0.1%, 0.0%) Nitrates; $n$ (%) 2,636 (4.2%) 3,482 (3.5%) 0.8% (0.6%, 1.0%) 1,196 (3.6%) 1,216 (3.7%) -0.1% (-0.3%, 0.2%) Anti-arrhythmics; $n$ (%) 881 (1.4%) 1,313 (1.3%) 0.1% (-0.6%, 0.2%) 432 (1.3%) 436 (1.3%) -0.0% (-0.2%, 0.2%) Statins; $n$ (%) 881 (1.4%) 1,313 (1.3%) 0.1% (-0.6%, 0.2%) 446 (1.3%) -0.0% (-0.2%, 0.2%) PCSK9 inhibitors and other lipid-lower | Past use of SGLT-2i; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ARNI; n (%) | 11,402 (18.3%)<br>4,351 (7.0%)<br>46,356 (74.2%)<br>352 (0.6%) | 23,796 (23.6%)<br>5,580 (5.5%)<br>70,619 (70.0%)<br>1,029 (1.0%) | -5.3% (-5.7%, -4.9%)<br>1.4% (1.2%, 1.7%)<br>4.2% (3.8%, 4.7%)<br>-0.5% (-0.5%, -0.4%) | 7,508 (22.6%)<br>2,242 (6.8%)<br>24,113 (72.7%)<br>221 (0.7%) | 7,761 (23.4%)<br>2,280 (6.9%)<br>24,155 (72.8%)<br>225 (0.7%) | -0.8% (-1.4%, -0.1%)<br>-0.1% (-0.5%, 0.3%)<br>-0.1% (-0.8%, 0.6%)<br>-0.0% (-0.1%, 0.1%) |
| Digoxin / Digitoxin; n (%) 366 (0.6%) 309 (0.3%) 0.3% (0.2%, 0.3%) 137 (0.4%) 136 (0.4%) 0.0% (-0.1%, 0.1%) Loop diuretics; n (%) 6,024 (9.6%) 9.811 (9.7%) -0.1% (-0.4%, 0.2%) 3,005 (9.1%) 3,016 (9.1%) -0.0% (-0.5%, 0.2%) Other diuretics; n (%) 3,731 (6.0%) 7,652 (7.6%) -1.6% (1.9%, 1.4%) 20.92 (6.3%) 2148 (6.5%) -0.2% (-0.5%, 0.2%) Intravenous diuretics; n (%) 331 (0.5%) 565 (0.6%) -0.0% (-0.1%, 0.0%) 153 (0.5%) 154 (0.5%) -0.0% (-0.1%, 0.0%) Nitrates; n (%) 2,636 (4.2%) 3,482 (3.5%) 0.8% (0.6%, 1.0%) 1,196 (3.6%) 1,216 (3.7%) -0.1% (-0.3%, 0.2%) Anti-arrhythmics; n (%) 881 (1.4%) 1,313 (1.3%) 0.1% (-0.0%, 0.2%) 432 (1.3%) 436 (1.3%) -0.0% (-0.2%, 0.2%) Statins; n (%) 46,719 (74.8%) 72,447 (71.8%) 3.0% (2.5%, 3.4%) 24,612 (74.2%) 24,647 (74.3%) -0.1% (-0.2%, 0.2%) Statins; n (%) 7,580 (12.1%) 11,487 (11.4%) 0.7% (0.4%, 1.1%) 3,925 (11.8%) 4,013 (12.1%) -0.3% (-0.8%, 0.2%) Oral anticoagulants; n (%) 6,224 (10.0%) 8,005 (7.9%) 2.0% (1.7%, 2.3%) 2,902 | Past use of SGLT-2i; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ARNI; n (%) Thiazides; n (%) | 11,402 (18.3%)<br>4,351 (7.0%)<br>46,356 (74.2%)<br>352 (0.6%)<br>20,945 (33.5%) | 23,796 (23.6%)<br>5,580 (5.5%)<br>70,619 (70.0%)<br>1,029 (1.0%)<br>35,859 (35.6%) | -5.3% (-5.7%, -4.9%)<br>1.4% (1.2%, 1.7%)<br>4.2% (3.8%, 4.7%)<br>-0.5% (-0.5%, -0.4%)<br>-2.0% (-2.5%, -1.5%) | 7,508 (22.6%)<br>2,242 (6.8%)<br>24,113 (72.7%)<br>221 (0.7%)<br>11,443 (34.5%) | 7,761 (23.4%)<br>2,280 (6.9%)<br>24,155 (72.8%)<br>225 (0.7%)<br>11,415 (34.4%) | -0.8% (-1.4%, -0.1%)<br>-0.1% (-0.5%, 0.3%)<br>-0.1% (-0.8%, 0.6%)<br>-0.0% (-0.1%, 0.1%)<br>0.1% (-0.6%, 0.8%) |
| Loop diuretics; n (%) 6,024 (9.6%) 9,811 (9.7%) -0.1% (-0.4%, 0.2%) 3,005 (9.1%) 3,016 (9.1%) -0.0% (-0.5%, 0.0) -0.0% (-0.5%, | Past use of SGLT-2i; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ARNI; n (%) Thiazides; n (%) Beta-blockers; n (%) | 11,402 (18.3%)<br>4,351 (7.0%)<br>46,356 (74.2%)<br>352 (0.6%)<br>20,945 (33.5%)<br>20,935 (33.5%) | 23,796 (23.6%)<br>5,580 (5.5%)<br>70,619 (70.0%)<br>1,029 (1.0%)<br>35,859 (35.6%)<br>31,879 (31.6%) | -5.3% (-5.7%, -4.9%)<br>1.4% (1.2%, 1.7%)<br>4.2% (3.8%, 4.7%)<br>-0.5% (-0.5%, -0.4%)<br>-2.0% (-2.5%, -1.5%)<br>1.9% (1.4%, 2.4%) | 7,508 (22.6%)<br>2,242 (6.8%)<br>24,113 (72.7%)<br>221 (0.7%)<br>11,443 (34.5%)<br>10,504 (31.6%) | 7,761 (23.4%)<br>2,280 (6.9%)<br>24,155 (72.8%)<br>225 (0.7%)<br>11,415 (34.4%)<br>10,528 (31.7%) | -0.8% (-1.4%, -0.1%)<br>-0.1% (-0.5%, 0.3%)<br>-0.1% (-0.8%, 0.6%)<br>-0.0% (-0.1%, 0.1%)<br>0.1% (-0.6%, 0.8%)<br>-0.1% (-0.8%, 0.6%) |
| Other diuretics; n (%) 3,731 (6.0%) 7,652 (7.6%) -1.6% (-1.9%, -1.4%) 2.092 (6.3%) 2,148 (6.5%) -0.2% (-0.5%, 0.2%) Intravenous diuretics; n (%) 331 (0.5%) 565 (0.6%) -0.0% (-0.1%, 0.0%) 153 (0.5%) 154 (0.5%) -0.0% (-0.1%, 0.1%) Nitrates; n (%) 2,636 (4.2%) 3,482 (3.5%) 0.8% (0.6%, 1.0%) 1,196 (3.6%) 1,216 (3.7%) -0.1% (-0.3%, 0.2%) Anti-arrhythmics; n (%) 881 (1.4%) 1,313 (1.3%) 0.1% (-0.0%, 0.2%) 432 (1.3%) 436 (1.3%) -0.0% (-0.2%, 0.2%) Statins; n (%) 46,719 (74.8%) 72,447 (71.8%) 3.0% (2.5%, 3.4%) 24,612 (74.2%) 24,647 (74.3%) -0.0% (-0.8%, 0.2%) PCSK9 inhibitors and other lipid-lowering drugs; n (%) 7,580 (12.1%) 11,487 (11.4%) 0.7% (0.4%, 11%) 3,925 (11.8%) 4,013 (12.1%) -0.3% (-0.8%, 0.2%) Antiplatelet medications; n (%) 6,224 (10.0%) 8,005 (7.9%) 2.0% (1.7%, 2.3%) 2,902 (8.7%) 2,967 (8.9%) 0.2% (-0.6%, 0.2%) Oral anticoagulants; n (%) 4,068 (6.5%) 5,754 (5.7%) 0.8% (0.6%, 11%) 1,940 (5.8%) 1,957 (5.9%) -0.1% (-0.4%, 0.3 <td>Past use of SGLT-2i; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ARNI; n (%) Thiazides; n (%) Beta-blockers; n (%) Calcium channel blockers; n (%)</td> <td>11,402 (18.3%)<br/>4,351 (7.0%)<br/>46,356 (74.2%)<br/>352 (0.6%)<br/>20,945 (33.5%)<br/>20,935 (33.5%)<br/>18,193 (29.1%)</td> <td>23,796 (23.6%)<br/>5,580 (5.5%)<br/>70,619 (70.0%)<br/>1,029 (1.0%)<br/>35,859 (35.6%)<br/>31,879 (31.6%)<br/>27,539 (27.3%)</td> <td>-5.3% (-5.7%, -4.9%)<br/>1.4% (1.2%, 1.7%)<br/>4.2% (3.8%, 4.7%)<br/>-0.5% (-0.5%, -0.4%)<br/>-2.0% (-2.5%, -1.5%)<br/>1.9% (1.4%, 2.4%)<br/>1.8% (1.4%, 2.3%)</td> <td>7,508 (22.6%)<br/>2,242 (6.8%)<br/>24,113 (72.7%)<br/>221 (0.7%)<br/>11,443 (34.5%)<br/>10,504 (31.6%)<br/>9,267 (27.9%)</td> <td>7,761 (23.4%)<br/>2,280 (6.9%)<br/>24,155 (72.8%)<br/>225 (0.7%)<br/>11,415 (34.4%)<br/>10,528 (31.7%)<br/>9,183 (27.7%)</td> <td>-0.8% (-1.4%, -0.1%)<br/>-0.1% (-0.5%, 0.3%)<br/>-0.1% (-0.8%, 0.6%)<br/>-0.0% (-0.1%, 0.1%)<br/>-0.0% (-0.6%, 0.8%)<br/>-0.1% (-0.8%, 0.6%)<br/>0.3% (-0.4%, 0.9%)</td> | Past use of SGLT-2i; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ARNI; n (%) Thiazides; n (%) Beta-blockers; n (%) Calcium channel blockers; n (%) | 11,402 (18.3%)<br>4,351 (7.0%)<br>46,356 (74.2%)<br>352 (0.6%)<br>20,945 (33.5%)<br>20,935 (33.5%)<br>18,193 (29.1%) | 23,796 (23.6%)<br>5,580 (5.5%)<br>70,619 (70.0%)<br>1,029 (1.0%)<br>35,859 (35.6%)<br>31,879 (31.6%)<br>27,539 (27.3%) | -5.3% (-5.7%, -4.9%)<br>1.4% (1.2%, 1.7%)<br>4.2% (3.8%, 4.7%)<br>-0.5% (-0.5%, -0.4%)<br>-2.0% (-2.5%, -1.5%)<br>1.9% (1.4%, 2.4%)<br>1.8% (1.4%, 2.3%) | 7,508 (22.6%)<br>2,242 (6.8%)<br>24,113 (72.7%)<br>221 (0.7%)<br>11,443 (34.5%)<br>10,504 (31.6%)<br>9,267 (27.9%) | 7,761 (23.4%)<br>2,280 (6.9%)<br>24,155 (72.8%)<br>225 (0.7%)<br>11,415 (34.4%)<br>10,528 (31.7%)<br>9,183 (27.7%) | -0.8% (-1.4%, -0.1%)<br>-0.1% (-0.5%, 0.3%)<br>-0.1% (-0.8%, 0.6%)<br>-0.0% (-0.1%, 0.1%)<br>-0.0% (-0.6%, 0.8%)<br>-0.1% (-0.8%, 0.6%)<br>0.3% (-0.4%, 0.9%) |
| $ \begin{array}{c ccccccccccccccccccccccccccccccccccc$ | Past use of SGLT-2i; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ARNI; n (%) Thiazides; n (%) Beta-blockers; n (%) Calcium channel blockers; n (%) Digoxin / Digitoxin; n (%) | 11,402 (18.3%) 4,351 (7.0%) 46,356 (74.2%) 352 (0.6%) 20,945 (33.5%) 20,935 (33.5%) 18,193 (29.1%) 366 (0.6%) | 23,796 (23.6%)<br>5,580 (5.5%)<br>70,619 (70.0%)<br>1,029 (1.0%)<br>35,859 (35.6%)<br>31,879 (31.6%)<br>27,539 (27.3%)<br>309 (0.3%) | -5.3% (-5.7%, -4.9%)<br>1.4% (1.2%, 1.7%)<br>4.2% (3.8%, 4.7%)<br>-0.5% (-0.5%, -0.4%)<br>-2.0% (-2.5%, -1.5%)<br>1.9% (1.4%, 2.4%)<br>1.8% (1.4%, 2.3%)<br>0.3% (0.2%, 0.3%) | 7,508 (22.6%)<br>2,242 (6.8%)<br>24,113 (72.7%)<br>221 (0.7%)<br>11,443 (34.5%)<br>10,504 (31.6%)<br>9,267 (27.9%)<br>137 (0.4%) | 7,761 (23.4%)<br>2,280 (6.9%)<br>24,155 (72.8%)<br>225 (0.7%)<br>11,415 (34.4%)<br>10,528 (31.7%)<br>9,183 (27.7%)<br>136 (0.4%) | -0.8% (-1.4%, -0.1%)<br>-0.1% (-0.5%, 0.3%)<br>-0.1% (-0.8%, 0.6%)<br>-0.0% (-0.1%, 0.1%)<br>-0.1% (-0.6%, 0.8%)<br>-0.1% (-0.6%, 0.6%)<br>-0.3% (-0.4%, 0.9%)<br>-0.0% (-0.1%, 0.1%) |
| Nitrates; $n$ (%) 2.636 (4.2%) 3.482 (3.5%) 0.8% (0.6%, 1.0%) 1.196 (3.6%) 1.216 (3.7%) -0.1% (-0.3%, 0.2 Anti-arrhythmics; $n$ (%) 881 (1.4%) 1.313 (1.3%) 0.1% (-0.0%, 0.2%) 432 (1.3%) 436 (1.3%) -0.0% (-0.2%, 0.2 Statins; $n$ (%) 46,719 (74.8%) 72,447 (71.8%) 3.0% (2.5%, 3.4%) 24,612 (74.2%) 24,647 (74.3%) -0.1% (-0.8%, 0.2 Anti-plate in medications; $n$ (%) 7.580 (12.1%) 11,487 (11.4%) 0.7% (0.4%, 1.1%) 3.925 (11.8%) 4.013 (12.1%) -0.3% (-0.8%, 0.2 Anti-plate in medications; $n$ (%) 6,224 (10.0%) 8,005 (7.9%) 2.0% (1.7%, 2.3%) 2.902 (8.7%) 2.967 (8.9%) -0.2% (-0.6%, 0.2 Anti-plate in medications; $n$ (%) 4,068 (6.5%) 5,754 (5.7%) 0.8% (0.6%, 1.1%) 1.940 (5.8%) 1.957 (5.9%) 0.1% (-0.4%, 0.2 COPD/Asthma medications; $n$ (%) 17,438 (27.9%) 32,810 (32.5%) -4.6% (-5.1%, -4.2%) 9,768 (29.4%) 1.957 (3.9%) 0.1% (-0.4%, 0.2 COPD/Asthma medications; $n$ (%) 19,570 (3.3%) 34,820 (34.5%) 3.2% (3.3%, 2.7%) 10,961 (33.0%) 10,910 (32.9%) 0.2% (-0.6%, 0.2 COPD/Asthma medications; $n$ (%) 12,920 (20.7%) 26,471 (26.2%) -5.6% (-6.0%, 5.1%) 7,444 (22.4%) 7,345 (22.1%) 0.3% (-0.3%, 0.5 COPD/Asthma medications; $n$ (%) 12,920 (20.7%) 26,471 (26.2%) -5.6% (-6.0%, 5.1%) 7,444 (22.4%) 7,345 (22.1%) 0.3% (-0.3%, 0.5 COPD/Asthma medications; $n$ (%) 12,920 (20.7%) 26,471 (26.2%) -5.6% (-6.0%, 5.1%) 7,444 (22.4%) 7,345 (22.1%) 0.3% (-0.3%, 0.5 COPD/Asthma medications; $n$ (%) 12,920 (20.7%) 26,471 (26.2%) -5.6% (-6.0%, 5.1%) 7,444 (22.4%) 7,345 (22.1%) 0.3% (-0.3%, 0.5 COPD/Asthma medications; $n$ (%) 12,920 (20.7%) 26,471 (26.2%) -5.6% (-6.0%, 5.1%) 7,444 (22.4%) 7,345 (22.1%) 0.3% (-0.3%, 0.5 COPD/Asthma medications; $n$ (%) 12,920 (20.7%) 26,471 (26.2%) -5.6% (-6.0%, 5.1%) 7,444 (22.4%) 7,345 (22.1%) 0.3% (-0.3%, 0.5 COPD/Asthma medications; $n$ (%) 12,920 (20.7%) 26,471 (26.2%) -5.6% (-6.0%, 5.1%) 7,444 (22.4%) 7,345 (22.1%) 0.3% (-0.3%, 0.5 COPD/Asthma medications; $n$ (%) 12,920 (20.7%) 26,471 (26.2%) -5.6% (-6.0%, 5.1%) 7,444 (22.4%) 7,345 (22.1%) 0.3% (-0.3%, 0.5 COPD/Asthma medications; $n$ (%) 12,920 (20.7%) 26,471 (26.2%) 1 | Past use of SGLT-2i; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ARNI; n (%) Thiazides; n (%) Beta-blockers; n (%) Calcium channel blockers; n (%) Digoxin / Digitoxin; n (%) Loop diuretics; n (%) | 11,402 (18.3%) 4,351 (7.0%) 46,356 (74.2%) 352 (0.6%) 20,945 (33.5%) 20,935 (33.5%) 18,193 (29.1%) 366 (0.6%) 6,024 (9.6%) | 23,796 (23.6%) 5,580 (5.5%) 70,619 (70.0%) 1,029 (10%) 35,859 (35.6%) 31,879 (31.6%) 27,539 (27.3%) 309 (0.3%) 9,811 (9.7%) | -5.3% (-5.7%, -4.9%)<br>1.4% (1.2%, 1.7%)<br>4.2% (3.8%, 4.7%)<br>-0.5% (-0.5%, -0.4%)<br>-2.0% (-2.5%, -1.5%)<br>1.9% (1.4%, 2.4%)<br>1.8% (1.4%, 2.3%)<br>-0.3% (0.2%, 0.3%)<br>-0.1% (-0.4%, 0.2%) | 7.508 (22.6%)<br>2.242 (6.8%)<br>24,113 (72.7%)<br>221 (0.7%)<br>11,443 (34.5%)<br>10,504 (31.6%)<br>9,504 (31.6%)<br>137 (0.4%)<br>3,005 (9.1%) | 7.761 (23.4%)<br>2.280 (6.9%)<br>24,155 (72.8%)<br>225 (0.7%)<br>11,415 (34.4%)<br>10,528 (31.7%)<br>9,183 (27.7%)<br>136 (0.4%)<br>3,016 (9.1%) | -0.8% (-1.4%, -0.1%)<br>-0.1% (-0.5%, 0.3%)<br>-0.1% (-0.8%, 0.6%)<br>-0.0% (-0.1%, 0.1%)<br>0.1% (-0.6%, 0.8%)<br>-0.1% (-0.8%, 0.6%)<br>0.3% (-0.4%, 0.9%)<br>-0.0% (-0.1%, 0.1%)<br>-0.0% (-0.1%, 0.1%) |
| $ \begin{array}{cccccccccccccccccccccccccccccccccccc$ | Past use of SGLT-2i; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ARNI; n (%) Thiazides; n (%) Beta-blockers; n (%) Calcium channel blockers; n (%) Digoxin / Digitoxin; n (%) Loop diuretics; n (%) Other diuretics; n (%) | 11,402 (18.3%) 4,351 (7.0%) 46,356 (74.2%) 352 (0.6%) 20,945 (33.5%) 20,935 (33.5%) 18,193 (29.1%) 366 (0.6%) 6,024 (9.6%) 3,731 (6.0%) | 23,796 (23.6%) 5,580 (5.5%) 70,619 (70.0%) 1,029 (1.0%) 35,859 (35.6%) 31,879 (31.6%) 27,539 (27.3%) 309 (0.3%) 9,811 (9.7%) 7,652 (7.6%) | -5.3% (-5.7%, -4.9%)<br>1.4% (1.2%, 1.7%)<br>4.2% (3.8%, 4.7%)<br>-0.5% (-0.5%, -0.4%)<br>-2.0% (-2.5%, -1.5%)<br>1.9% (1.4%, 2.4%)<br>1.8% (1.4%, 2.3%)<br>0.3% (0.2%, 0.3%)<br>-0.1% (-0.4%, 0.2%)<br>-1.6% (-1.9%, -1.4%) | 7.508 (22.6%) 2.242 (6.8%) 24,113 (72.7%) 221 (0.7%) 11,443 (34.5%) 10,504 (31.6%) 9,267 (27.9%) 137 (0.4%) 3,005 (9.1%) 2,092 (6.3%) | 7,761 (23.4%)<br>2,280 (6.9%)<br>24,155 (72.8%)<br>225 (0.7%)<br>11,415 (34.4%)<br>10,528 (31.7%)<br>9,183 (27.7%)<br>136 (0.4%)<br>3,016 (9.1%)<br>2,148 (6.5%) | -0.8% (-1.4%, -0.1%)<br>-0.1% (-0.5%, 0.3%)<br>-0.1% (-0.5%, 0.6%)<br>-0.0% (-0.1%, 0.1%)<br>-0.1% (-0.8%, 0.6%)<br>-0.1% (-0.8%, 0.6%)<br>-0.3% (-0.4%, 0.9%)<br>-0.0% (-0.1%, 0.1%)<br>-0.0% (-0.5%, 0.4%)<br>-0.2% (-0.5%, 0.2%) |
| $ \begin{array}{cccccccccccccccccccccccccccccccccccc$ | Past use of SGLT-2i; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ARNI; n (%) Thiazides; n (%) Beta-blockers; n (%) Calcium channel blockers; n (%) Digoxin / Digitoxin; n (%) Loop diuretics; n (%) Other diuretics; n (%) Intravenous diuretics; n (%) | 11,402 (18.3%) 4.351 (7.0%) 46,356 (74.2%) 352 (0.6%) 20,945 (33.5%) 20,935 (33.5%) 18,193 (29.1%) 366 (0.6%) 6,024 (9.6%) 3,731 (6.0%) 331 (0.5%) | 23,796 (23.6%) 5,580 (5.5%) 70,619 (70.0%) 1,029 (1.0%) 35,859 (35.6%) 31,879 (31.6%) 27,539 (27.3%) 309 (0.3%) 9,811 (9.7%) 7,652 (7.6%) 565 (0.6%) | -5.3% (-5.7%, -4.9%)<br>1.4% (1.2%, 1.7%)<br>4.2% (3.8%, 4.7%)<br>-0.5% (-0.5%, -0.4%)<br>-2.0% (-2.5%, -1.5%)<br>1.9% (1.4%, 2.4%)<br>1.8% (1.4%, 2.3%)<br>0.3% (0.2%, 0.3%)<br>-0.1% (-0.4%, 0.2%)<br>-1.6% (-1.9%, -1.4%)<br>-0.0% (-0.1%, 0.0%) | 7,508 (22.6%) 2,242 (6.8%) 24,113 (72.7%) 24,113 (72.7%) 11,443 (34.5%) 10,504 (31.6%) 9,267 (27.9%) 137 (0.4%) 3,005 (9.1%) 2,092 (6.3%) 153 (0.5%) | 7,761 (23.4%)<br>2,280 (6.9%)<br>24,155 (72.8%)<br>225 (0.7%)<br>11,415 (34.4%)<br>10,528 (31.7%)<br>9,183 (27.7%)<br>136 (0.4%)<br>3,016 (9.1%)<br>2,148 (6.5%)<br>154 (0.5%) | -0.8% (-1.4%, -0.1%)<br>-0.1% (-0.5%, 0.3%)<br>-0.1% (-0.8%, 0.6%)<br>-0.0% (-0.1%, 0.1%)<br>-0.1% (-0.6%, 0.8%)<br>-0.1% (-0.6%, 0.8%)<br>-0.1% (-0.4%, 0.9%)<br>-0.0% (-0.1%, 0.1%)<br>-0.0% (-0.5%, 0.4%)<br>-0.2% (-0.5%, 0.2%)<br>-0.0% (-0.1%, 0.1%) |
| $ \begin{array}{cccccccccccccccccccccccccccccccccccc$ | Past use of SGLT-2i; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ARNI; n (%) Thiazides; n (%) Beta-blockers; n (%) Digoxin / Digitoxin; n (%) Loop diuretics; n (%) Other diuretics; n (%) Intravenous diuretics; n (%) Nitrates; n (%) | 11,402 (18.3%) 4,351 (7.0%) 46,356 (74.2%) 352 (0.6%) 20,945 (33.5%) 20,935 (33.5%) 18,193 (29.1%) 366 (0.6%) 6,024 (9.6%) 3,731 (6.0%) 331 (0.5%) 2,636 (4.2%) | 23,796 (23.6%) 5,580 (5.5%) 70,619 (70.0%) 1,029 (1.0%) 35,859 (35.6%) 31,879 (31.6%) 27,539 (27.3%) 309 (0.3%) 9,811 (9.7%) 7,652 (7.6%) 565 (0.6%) 3,482 (3.5%) | -5.3% (-5.7%, -4.9%)<br>1.4% (1.2%, 1.7%)<br>4.2% (3.8%, 4.7%)<br>-0.5% (-0.5%, -0.4%)<br>-2.0% (-2.5%, -1.5%)<br>1.9% (1.4%, 2.3%)<br>0.3% (0.2%, 0.3%)<br>-0.1% (-0.4%, 0.2%)<br>-1.6% (-1.9%, -1.4%)<br>-0.0% (-0.1%, 0.0%)<br>0.8% (0.6%, 1.0%) | 7,508 (22.6%) 2,242 (6.8%) 2,413 (72.7%) 221 (0.7%) 11,443 (34.5%) 10,504 (31.6%) 9,267 (27.9%) 137 (0.4%) 3,005 (9.1%) 2,002 (6.3%) 153 (0.5%) 1,196 (3.6%) | 7,761 (23.4%) 2,280 (6.9%) 24,155 (72.8%) 225 (0.7%) 11,415 (34.4%) 10,528 (31.7%) 136 (0.4%) 3,016 (9.1%) 2,148 (6.5%) 154 (0.5%) 1,216 (3.7%) | -0.8% (-1.4%, -0.1%) -0.1% (-0.5%, 0.3%) -0.1% (-0.5%, 0.3%) -0.0% (-0.1%, 0.1%) -0.1% (-0.6%, 0.8%) -0.1% (-0.6%, 0.9%) -0.1% (-0.6%, 0.9%) -0.0% (-0.1%, 0.1%) -0.0% (-0.1%, 0.1%) -0.0% (-0.5%, 0.4%) -0.2% (-0.5%, 0.2%) -0.0% (-0.1%, 0.1%) -0.0% (-0.1%, 0.1%) |
| Antiplatelet medications; n (%) 6,224 (10.0%) 8,005 (7.9%) 2.0% (1.7%, 2.3%) 2,902 (8.7%) 2,967 (8.9%) -0.2% (-0.6%, 0.2%) -0. | Past use of SGLT-2i; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ARNI; n (%) Thiazides; n (%) Beta-blockers; n (%) Calcium channel blockers; n (%) Digoxin / Digitoxin; n (%) Loop diuretics; n (%) Other diuretics; n (%) Intravenous diuretics; n (%) Nitrates; n (%) Anti-arrhythmics; n (%) | 11,402 (18.3%) 4,351 (7.0%) 46,356 (74.2%) 352 (0.6%) 20,945 (33.5%) 20,935 (33.5%) 18,193 (29.1%) 366 (0.6%) 6,024 (9.6%) 3,731 (6.0%) 331 (0.5%) 2,636 (4.2%) 881 (1.4%) | 23,796 (23.6%) 5,580 (5.5%) 70,619 (70.0%) 1,029 (10%) 35,859 (35.6%) 31,879 (31.6%) 27,539 (27.3%) 309 (0.3%) 9,811 (9.7%) 7,652 (7.6%) 565 (0.6%) 3,482 (3.5%) 1,313 (1.3%) | -5.3% (-5.7%, -4.9%)<br>1.4% (1.2%, 1.7%)<br>4.2% (3.8%, 4.7%)<br>-0.5% (-0.5%, -0.4%)<br>-2.0% (-2.5%, -1.5%)<br>1.9% (1.4%, 2.4%)<br>1.8% (1.4%, 2.3%)<br>-0.3% (0.2%, 0.3%)<br>-0.1% (-0.4%, 0.2%)<br>-1.6% (-1.9%, -1.4%)<br>-0.0% (-0.1%, 0.0%)<br>0.3% (0.5%, 1.0%) | 7,508 (22.6%) 2,242 (6.8%) 2,413 (72.7%) 221 (0.7%) 11,443 (34.5%) 10,504 (31.6%) 9,267 (27.9%) 137 (0.4%) 3,005 (9.1%) 2,092 (6.3%) 153 (0.5%) 1,196 (3.6%) 432 (1.3%) | 7,761 (23.4%) 2,280 (6.9%) 2,4,155 (72.8%) 225 (0.7%) 11,415 (34.4%) 10,528 (31.7%) 136 (0.4%) 3,016 (9.1%) 2,148 (6.5%) 154 (0.5%) 1,216 (3.7%) 436 (1.3%) | -0.8% (-1.4%, -0.1%) -0.1% (-0.5%, 0.3%) -0.1% (-0.5%, 0.3%) -0.1% (-0.8%, 0.6%) -0.0% (-0.1%, 0.1%) 0.1% (-0.6%, 0.8%) -0.1% (-0.8%, 0.6%) 0.3% (-0.4%, 0.9%) -0.0% (-0.1%, 0.1%) -0.0% (-0.5%, 0.4%) -0.2% (-0.5%, 0.2%) -0.0% (-0.1%, 0.1%) -0.0% (-0.1%, 0.1%) -0.0% (-0.0%, 0.2%) -0.0% (-0.3%, 0.2%) |
| $ \begin{array}{cccccccccccccccccccccccccccccccccccc$ | Past use of SGLT-2i; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ARNI; n (%) Thiazides; n (%) Beta-blockers; n (%) Calcium channel blockers; n (%) Digoxin / Digitoxin; n (%) Loop diuretics; n (%) Other diuretics; n (%) Intravenous diuretics; n (%) Nitrates; n (%) Statins; n (%) Statins; n (%) | 11,402 (18.3%) 4,351 (7.0%) 46,356 (74.2%) 352 (0.6%) 20,945 (33.5%) 20,935 (33.5%) 18,193 (29.1%) 366 (0.6%) 6,024 (9.6%) 3,731 (6.0%) 331 (0.5%) 2,636 (4.2%) 881 (4.4%) 46,719 (74.8%) | 23,796 (23.6%) 5,580 (5.5%) 70,619 (70.0%) 1,029 (1.0%) 35,859 (35.6%) 31,879 (31.6%) 27,539 (27.3%) 309 (0.3%) 9,811 (9.7%) 7,652 (7.6%) 565 (0.6%) 3,482 (3.5%) 1,313 (1.3%) 72,447 (71.8%) | -5.3% (-5.7%, -4.9%) 1.4% (1.2%, 1.7%) 4.2% (3.8%, 4.7%) 4.2% (3.8%, 4.7%) -0.5% (-0.5%, -0.4%) -2.0% (-2.5%, -1.5%) 1.9% (1.4%, 2.4%) 1.8% (1.4%, 2.3%) 0.3% (0.2%, 0.3%) -0.1% (-0.4%, 0.2%) -1.6% (-1.9%, -1.4%) -0.0% (-0.1%, 0.0%) 0.1% (-0.0%, 0.0%) 0.1% (-0.0%, 0.0%) | 7.508 (22.6%) 2.242 (6.8%) 2.4113 (72.7%) 221 (0.7%) 11,443 (34.5%) 10,504 (31.6%) 9.267 (27.9%) 137 (0.4%) 3.005 (9.1%) 2.092 (6.3%) 153 (0.5%) 1,196 (3.6%) 432 (1.3%) 24,612 (74.2%) | 7,761 (23.4%) 2,280 (6.9%) 24,155 (72.8%) 225 (0.7%) 11,415 (34.4%) 10,528 (31.7%) 9,183 (27.7%) 136 (0.4%) 3,016 (91%) 2,148 (6.5%) 154 (0.5%) 152 (3.7%) 436 (1.3%) 436 (1.3%) 24,647 (74.3%) | -0.8% (-1.4%, -0.1%) -0.1% (-0.5%, 0.3%) -0.1% (-0.5%, 0.3%) -0.1% (-0.8%, 0.6%) -0.0% (-0.1%, 0.1%) -0.1% (-0.8%, 0.6%) -0.3% (-0.4%, 0.9%) -0.0% (-0.1%, 0.1%) -0.0% (-0.5%, 0.4%) -0.2% (-0.5%, 0.2%) -0.0% (-0.1%, 0.1%) -0.1% (-0.3%, 0.2%) -0.0% (-0.2%, 0.2%) -0.1% (-0.3%, 0.2%) -0.1% (-0.3%, 0.2%) |
| $ \begin{array}{cccccccccccccccccccccccccccccccccccc$ | Past use of SGLT-2i; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ACE-is/ARB's; n (%) Beta-blockers; n (%) Beta-blockers; n (%) Calcium channel blockers; n (%) Digoxin / Digitoxin; n (%) Loop diuretics; n (%) Other diuretics; n (%) Intravenous diuretics; n (%) Nitrates; n (%) Anti-arrhythmics; n (%) Statins; n (%) PCSK9 inhibitors and other lipid-lowering drugs; n (%) | 11,402 (18.3%) 4,351 (7.0%) 46,356 (74.2%) 352 (0.6%) 20,945 (33.5%) 20,935 (33.5%) 18,193 (29.1%) 366 (0.6%) 6,024 (9.6%) 3,731 (6.0%) 3,311 (0.5%) 2,636 (4.2%) 881 (1.4%) 46,719 (74.8%) 7,580 (12.1%) | 23,796 (23.6%) 5,580 (5.5%) 70,619 (70.0%) 1,029 (1.0%) 35,859 (35.6%) 31,879 (31.6%) 27,539 (27.3%) 309 (0.3%) 9,811 (9.7%) 7,652 (7.6%) 565 (0.6%) 3,482 (3.5%) 1,313 (1.3%) 1,2447 (71.8%) 11,487 (11.4%) | -5.3% (-5.7%, -4.9%) 1.4% (1.2%, 1.7%) 4.2% (3.8%, 4.7%) -0.5% (-0.5%, -0.4%) -2.0% (-2.5%, -1.5%) 1.9% (1.4%, 2.4%) 1.8% (1.4%, 2.3%) 0.3% (0.2%, 0.3%) -0.1% (-0.4%, 0.2%) -1.6% (-1.9%, -1.4%) -0.0% (-0.1%, 0.0%) 0.8% (0.6%, 1.0%) 0.8% (0.6%, 1.0%) 0.3% (0.2%) 3.0% (2.25%, 3.4%) | 7,508 (22.6%) 2,242 (6.8%) 2,242 (6.8%) 24,113 (72.7%) 221 (0.7%) 11,443 (34.5%) 10,504 (31.6%) 9,267 (27.9%) 137 (0.4%) 3,005 (9.1%) 2,092 (6.3%) 153 (0.5%) 1,196 (3.6%) 432 (1.3%) 432 (1.3%) 3,925 (11.8%) | 7,761 (23.4%) 2,280 (6.9%) 24,155 (72.8%) 225 (0.7%) 11,415 (34.4%) 10,528 (31.7%) 136 (0.4%) 3,016 (9.1%) 154 (0.5%) 154 (0.5%) 1,216 (3.7%) 436 (1.3%) 436 (1.3%) 4,013 (12.1%) | -0.8% (-1.4%, -0.1%) -0.1% (-0.5%, 0.3%) -0.1% (-0.5%, 0.3%) -0.1% (-0.8%, 0.6%) -0.1% (-0.1%, 0.1%) -0.1% (-0.8%, 0.6%) -0.3% (-0.4%, 0.9%) -0.0% (-0.1%, 0.1%) -0.0% (-0.5%, 0.4%) -0.2% (-0.5%, 0.2%) -0.0% (-0.1%, 0.1%) -0.1% (-0.3%, 0.2%) -0.0% (-0.1%, 0.1%) -0.1% (-0.3%, 0.2%) -0.0% (-0.1%, 0.1%) |
| $ \begin{array}{cccccccccccccccccccccccccccccccccccc$ | Past use of SGLT-2i; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ARNI; n (%) Thiazides; n (%) Beta-blockers; n (%) Beta-blockers; n (%) Digoxin / Digitoxin; n (%) Loop diuretics; n (%) Other diuretics; n (%) Intravenous diuretics; n (%) Nitrates; n (%) Anti-arrhythmics; n (%) Statins; n (%) PCSK9 inhibitors and other lipid-lowering drugs; n (%) Antiplatelet medications; n (%) | 11,402 (18.3%) 4,351 (7.0%) 46,356 (74.2%) 352 (0.6%) 20,945 (33.5%) 20,935 (33.5%) 18,193 (29.1%) 366 (0.6%) 6,024 (9.6%) 3,731 (6.0%) 26,36 (4.2%) 881 (1.4%) 46,719 (74.8%) 7,580 (12.1%) 6,224 (10.0%) | 23,796 (23.6%) 5,580 (5.5%) 70,619 (70.0%) 1,029 (10%) 35,859 (35.6%) 31,879 (31.6%) 27,539 (27.3%) 309 (0.3%) 9,811 (9.7%) 7,652 (7.6%) 565 (0.6%) 3,482 (3.5%) 1,313 (1.3%) 72,447 (71.8%) 11,487 (11.4%) 8,005 (7.9%) | -5.3% (-5.7%, -4.9%) 1.4% (1.2%, 1.7%) 4.2% (3.8%, 4.7%) -0.5% (-0.5%, -0.4%) -2.0% (-2.5%, -1.5%) 1.9% (1.4%, 2.3%) 0.3% (0.2%, 0.3%) -0.1% (-0.4%, 0.2%) -1.6% (-1.9%, -1.4%) -0.0% (-0.1%, 0.0%) 0.8% (0.6%, 1.0%) 0.3% (0.2%, 0.3%) | 7,508 (22.6%) 2,242 (6.8%) 2,242 (6.8%) 24,113 (72.7%) 221 (0.7%) 11,443 (34.5%) 10,504 (31.6%) 9,267 (27.9%) 137 (0.4%) 3,005 (9.1%) 2,092 (6.3%) 1,196 (3.6%) 432 (1.3%) 24,612 (74.2%) 3,925 (11.8%) 2,902 (8.7%) | 7,761 (23.4%) 2,280 (6.9%) 2,4,155 (72.8%) 225 (0.7%) 11,415 (34.4%) 10,528 (31.7%) 9,183 (27.7%) 136 (0.4%) 3,016 (9.1%) 2,148 (6.5%) 1,216 (3.7%) 436 (1.3%) 24,647 (74.3%) 4,013 (12.1%) 2,967 (8.9%) | -0.8% (-1.4%, -0.1%) -0.1% (-0.5%, 0.3%) -0.1% (-0.5%, 0.3%) -0.0% (-0.1%, 0.1%) -0.1% (-0.6%, 0.8%) -0.1% (-0.6%, 0.8%) -0.1% (-0.6%, 0.9%) -0.3% (-0.4%, 0.9%) -0.0% (-0.1%, 0.1%) -0.0% (-0.1%, 0.1%) -0.0% (-0.5%, 0.4%) -0.2% (-0.5%, 0.2%) -0.0% (-0.2%, 0.2%) -0.0% (-0.2%, 0.2%) -0.0% (-0.2%, 0.2%) -0.1% (-0.3%, 0.6%) -0.3% (-0.8%, 0.6%) -0.3% (-0.8%, 0.6%) -0.3% (-0.0%, 0.2%) |
| Oral corticosteroids; n (%) 12,920 (20.7%) 26,471 (26.2%) -5.6% (-6.0%, -5.1%) 7,444 (22.4%) 7,345 (22.1%) 0.3% (-0.3%, 0.5.4%) | Past use of SGLT-2i; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ARNI; n (%) Thiazides; n (%) Beta-blockers; n (%) Beta-blockers; n (%) Calcium channel blockers; n (%) Digoxin / Digitoxin; n (%) Loop diuretics; n (%) Under diuretics; n (%) Intravenous diuretics; n (%) Intravenous diuretics; n (%) Anti-arrhythmics; n (%) Statins; n (%) PCSK9 inhibitors and other lipid-lowering drugs; n (%) Antiplatelet medications; n (%) Oral anticoagulants; n (%) | 11,402 (18.3%) 4,351 (7.0%) 46,356 (74.2%) 352 (0.6%) 20,945 (33.5%) 20,935 (33.5%) 18,193 (29.1%) 366 (0.6%) 6,024 (9.6%) 3,731 (6.0%) 331 (0.5%) 26,336 (4.2%) 881 (1.4%) 46,719 (74.8%) 7,580 (12.1%) 6,224 (10.0%) 4,068 (6.5%) | 23,796 (23.6%) 5,580 (5.5%) 70,619 (70.0%) 1,029 (10%) 35,859 (35.6%) 31,879 (31.6%) 27,539 (27.3%) 309 (0.3%) 9,811 (9.7%) 7,652 (7.6%) 565 (0.6%) 3,482 (3.5%) 1,313 (1.3%) 72,447 (71.8%) 11,487 (11.4%) 8,005 (7.9%) 5,754 (5.7%) | -5.3% (-5.7%, -4.9%) 1.4% (1.2%, 1.7%) 4.2% (3.8%, 4.7%) 4.2% (3.8%, 4.7%) -0.5% (-0.5%, -0.4%) -2.0% (-2.5%, -1.5%) 1.9% (1.4%, 2.4%) 1.8% (1.4%, 2.3%) -0.3% (0.2%, 0.3%) -0.1% (-0.4%, 0.2%) -1.6% (-1.9%, -1.4%) -0.0% (-0.1%, 0.0%) 0.1% (-0.0%, 0.2%) 3.0% (2.5%, 3.4%) 0.7% (0.4%, 1.1%) 2.0% (1.7%, 2.3%) 0.8% (0.6%, 1.1%) | 7.508 (22.6%) 2.242 (6.8%) 2.242 (6.8%) 2.413 (72.7%) 221 (0.7%) 11,443 (34.5%) 10,504 (31.6%) 9,267 (27.9%) 137 (0.4%) 3,005 (9.1%) 2.092 (6.3%) 153 (0.5%) 1,196 (3.6%) 432 (1.3%) 24,612 (74.2%) 3,925 (11.8%) 2.992 (8.7%) 1,940 (5.8%) | 7,761 (23.4%) 2,280 (6.9%) 24,155 (72.8%) 225 (0.7%) 11,415 (34.4%) 10,528 (31.7%) 136 (0.4%) 3,016 (9.1%) 2,148 (6.5%) 154 (0.5%) 1,216 (3.7%) 436 (1.3%) 4,013 (12.1%) 2,967 (8.9%) 1,957 (5.9%) | -0.8% (-1.4%, -0.1%) -0.1% (-0.5%, 0.3%) -0.1% (-0.5%, 0.3%) -0.1% (-0.8%, 0.6%) -0.0% (-0.1%, 0.1%) 0.1% (-0.6%, 0.8%) -0.1% (-0.8%, 0.6%) 0.3% (-0.4%, 0.9%) -0.0% (-0.1%, 0.1%) -0.0% (-0.1%, 0.1%) -0.0% (-0.5%, 0.2%) -0.0% (-0.1%, 0.1%) -0.1% (-0.3%, 0.2%) -0.1% (-0.4%, 0.3%) |
| | Past use of SGLT-2i; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ARNI; n (%) Thiazides; n (%) Beta-blockers; n (%) Calcium channel blockers; n (%) Digoxin / Digitoxin; n (%) Loop diuretics; n (%) Other diuretics; n (%) Intravenous diuretics; n (%) Nitrates; n (%) Anti-arrhythmics; n (%) Statins; n (%) PCSK9 inhibitors and other lipid-lowering drugs; n (%) Antiplatelet medications; n (%) Oral anticoagulants; n (%) Oral anticoagulants; n (%) | 11,402 (18.3%) 4,351 (7.0%) 46,356 (74.2%) 352 (0.6%) 20,945 (33.5%) 20,935 (33.5%) 18,193 (29.1%) 366 (0.6%) 6,024 (9.6%) 3,731 (6.0%) 331 (0.5%) 26,36 (4.2%) 881 (4.4%) 46,719 (74.8%) 7,580 (12.1%) 4,068 (6.5%) 17,438 (27.9%) | 23,796 (23.6%) 5,580 (5.5%) 70,619 (70.0%) 1,029 (10.0%) 35,859 (35.6%) 31,879 (31.6%) 27,539 (27.3%) 309 (0.3%) 9,811 (9.7%) 7,652 (7.6%) 565 (0.6%) 3,3482 (3.5%) 1,313 (1.3%) 72,447 (71.8%) 11,487 (11.4%) 8,005 (7.9%) 5,754 (5.7%) 32,810 (32.5%) | -5.3% (-5.7%, -4.9%) 1.4% (1.2%, 1.7%) 4.2% (3.8%, 4.7%) 4.2% (3.8%, 4.7%) -0.5% (-0.5%, -0.4%) -2.0% (-2.5%, -1.5%) 1.9% (1.4%, 2.4%) 1.8% (1.4%, 2.3%) -0.3% (0.2%, 0.3%) -0.1% (-0.4%, 0.2%) -1.6% (-1.9%, -1.4%) -0.0% (-0.1%, 0.0%) 0.8% (0.6%, 1.0%) 0.7% (0.4%, 0.1%) 3.0% (2.5%, 3.4%) 0.7% (0.4%, 1.1%) 2.0% (1.7%, 2.3%) 0.8% (0.6%, 1.1%) 4.6% (-5.1%, -4.2%) | 7.508 (22.6%) 2.242 (6.8%) 2.41.13 (72.7%) 221 (0.7%) 11,443 (34.5%) 10,504 (31.6%) 9.267 (27.9%) 3,005 (9.1%) 2.092 (6.3%) 153 (0.5%) 1,196 (3.6%) 432 (1.3%) 24,612 (74.2%) 3,925 (11.8%) 2,902 (8.7%) 1,940 (5.8%) 9,796 (29.5%) | 7,761 (23.4%) 2,280 (6.9%) 24,155 (72.8%) 225 (0.7%) 11,415 (34.4%) 10,528 (31.7%) 9,183 (27.7%) 3,016 (9.1%) 3,016 (9.1%) 1,216 (3.7%) 436 (1.3%) 4,013 (12.1%) 2,967 (8.9%) 1,957 (5.9%) 9,758 (29.4%) | -0.8% (-1.4%, -0.1%) -0.1% (-0.5%, 0.3%) -0.1% (-0.5%, 0.3%) -0.1% (-0.8%, 0.6%) -0.9% (-0.1%, 0.1%) 0.1% (-0.6%, 0.8%) -0.1% (-0.4%, 0.9%) 0.3% (-0.4%, 0.9%) -0.0% (-0.1%, 0.1%) -0.0% (-0.1%, 0.1%) -0.0% (-0.1%, 0.2%) -0.0% (-0.1%, 0.2%) -0.0% (-0.3%, 0.2%) -0.0% (-0.3%, 0.2%) -0.1% (-0.3%, 0.2%) -0.1% (-0.3%, 0.2%) -0.1% (-0.3%, 0.2%) -0.1% (-0.4%, 0.2%) -0.1% (-0.4%, 0.2%) -0.1% (-0.4%, 0.2%) |
| Osteoporosis agents (incl. bisphosphonates); n (%) 955 (1.5%) 1,196 (1.2%) 0.3% (0.2%, 0.5%) 431 (1.3%) 442 (1.3%) -0.0% (-0.2%, 0.5%) | Past use of SGLT-2i; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ARNI; n (%) Thiazides; n (%) Beta-blockers; n (%) Beta-blockers; n (%) Digoxin / Digitoxin; n (%) Loop diuretics; n (%) Other diuretics; n (%) Other diuretics; n (%) Nitrates; n (%) Nitrates; n (%) PCSK9 inhibitors and other lipid-lowering drugs; n (%) Anti-arrhythmics; n (%) Oral anticoagulants; n (%) Oral anticoagulants; n (%) COPD/Asthma medications; n (%) NSAIDS; n (%) | 11,402 (18.3%) 4,351 (7.0%) 4,351 (7.0%) 46,356 (74.2%) 352 (0.6%) 20,945 (33.5%) 20,935 (33.5%) 18,193 (29.1%) 366 (0.6%) 6,024 (9.6%) 3,731 (6.0%) 2,636 (4.2%) 881 (1.4%) 46,719 (74.8%) 7,580 (12.1%) 6,224 (10.0%) 4,068 (6.5%) 1,7438 (27.9%) 19,570 (31.3%) | 23,796 (23.6%) 5,580 (5.5%) 70,619 (70.0%) 1,029 (1.0%) 35,859 (35.6%) 31,879 (31.6%) 309 (0.3%) 309 (0.3%) 9,811 (9.7%) 7,652 (7.6%) 565 (0.6%) 3,482 (3.5%) 1,313 (1.3%) 1,2447 (71.8%) 11,487 (11.4%) 8,005 (7.9%) 5,754 (5.7%) 3,2810 (32.5%) 34,820 (34.5%) | -5.3% (-5.7%, -4.9%) 1.4% (1.2%, 1.7%) 4.2% (3.8%, 4.7%) -0.5% (-0.5%, -0.4%) -2.0% (-2.5%, -1.5%) 1.9% (1.4%, 2.4%) 1.8% (1.4%, 2.3%) 0.3% (0.2%, 0.3%) -0.1% (-0.4%, 0.2%) -1.6% (-1.9%, -1.4%) -0.0% (-0.1%, 0.0%) 0.8% (0.6%, 1.0%) 0.1% (-0.0%, 0.2%) 3.0% (2.5%, 3.4%) 0.7% (0.4%, 1.1%) 0.9% (0.4%, 1.1%) 0.9% (0.4%, 1.1%) 0.9% (0.6%, 1.1%) 0.8% (0.6%, 1.1%) 0.8% (0.6%, 1.1%) 0.8% (0.6%, 1.1%) 0.8% (0.6%, 1.1%) 0.8% (0.6%, 1.1%) | 7,508 (22.6%) 2,242 (6.8%) 2,242 (6.8%) 2,413 (72.7%) 221 (0.7%) 11,443 (34.5%) 10,504 (31.6%) 9,267 (27.9%) 137 (0.4%) 3,005 (9.1%) 2,092 (6.3%) 153 (0.5%) 1,196 (3.6%) 432 (1.3%) 432 (1.3%) 2,902 (8.7%) 1,940 (5.8%) 1,940 (5.8%) 1,940 (5.8%) 1,976 (29.5%) 10,961 (33.0%) | 7,761 (23.4%) 2,280 (6.9%) 2,4,155 (72.8%) 225 (0.7%) 11,415 (34.4%) 10,528 (31.7%) 136 (0.4%) 3,016 (9.1%) 1,54 (6.5%) 1,54 (6.5%) 1,216 (3.7%) 436 (1.3%) 436 (1.3%) 4,013 (12.1%) 2,967 (8.9%) 1,957 (5.9%) 1,975 (5.9%) 1,010 (32.9%) | -0.8% (-1.4%, -0.1%) -0.1% (-0.5%, 0.3%) -0.1% (-0.5%, 0.3%) -0.1% (-0.8%, 0.6%) -0.0% (-0.1%, 0.1%) -0.1% (-0.6%, 0.8%) -0.1% (-0.6%, 0.8%) -0.1% (-0.6%, 0.8%) -0.0% (-0.1%, 0.1%) -0.0% (-0.1%, 0.1%) -0.0% (-0.5%, 0.4%) -0.2% (-0.5%, 0.2%) -0.0% (-0.1%, 0.1%) -0.1% (-0.3%, 0.2%) -0.0% (-0.1%, 0.1%) -0.1% (-0.3%, 0.2%) -0.0% (-0.0%, 0.2%) -0.1% (-0.8%, 0.2%) -0.2% (-0.6%, 0.3%) -0.2% (-0.6%, 0.3%) -0.1% (-0.6%, 0.3%) |

| Opioids; n (%) | 16,005 (25.6%) | 26,257 (26.0%) | -0.4% (-0.8%, 0.0%) | 8,340 (25.1%) | 8,468 (25.5%) | -0.4% (-1.1%, 0.3%) |
|---|---|---|---|---|---|---|
| Anti-depressants; n (%) | 16,775 (26.9%) | 36,709 (36.4%) | -9.5% (-10.0%, -9.1%) | 10,111 (30.5%) | 10,178 (30.7%) | -0.2% (-0.9%, 0.5%) |
| Antipsychotics; n (%) | 1,492 (2.4%) | 2,981 (3.0%) | -0.6% (-0.7%, -0.4%) | 838 (2.5%) | 860 (2.6%) | -0.1% (-0.3%, 0.2%) |
| Anxiolytics / hypnotics, benzos; n (%) | 9,813 (15.7%) | 20,355 (20.2%) | -4.5% (-4.8%, -4.1%) | 5,743 (17.3%) | 5,682 (17.1%) | 0.2% (-0.4%, 0.8%) |
| Dementia medications; n (%) | 673 (1.1%) | 320 (0.3%) | 0.8% (0.7%, 0.8%) | 158 (0.5%) | 158 (0.5%) | 0.0% (-0.1%, 0.1%) |
| Urinary tract infections antibiotics; n (%) | 26,465 (42.4%) | 44,562 (44.2%) | -1.8% (-2.3%, -1.3%) | 14,049 (42.3%) | 14,162 (42.7%) | -0.3% (-1.1%, 0.4%) |
| Laxatives; n (%) | 1,550 (2.5%) | 2,946 (2.9%) | -0.4% (-0.6%, -0.3%) | 832 (2.5%) | 850 (2.6%) | -0.1% (-0.3%, 0.2%) |
| Number of distinct medications | | | | | | |
| mean (sd) | 11.96 (6.02) | 13.17 (6.44) | -1.21 (-1.27, -1.15) | 12.39 (6.31) | 12.46 (5.91) | -0.07 (-0.16, 0.03) |
| median [IQR] | 11.00 [8.00, 15.00] | 12.00 [9.00, 17.00] | - (-, -) | 11.00 [8.00, 16.00] | 11.00 [8.00, 16.00] | - (-, -) |
| min, max | 1.00, 66.00 | 1.00, 72.00 | - (-, -) | 1.00, 66.00 | 1.00, 62.00 | - (-, -) |
| Number of office visits | | | | | | |
| mean (sd) | 7.61 (5.98) | 8.40 (6.30) | -0.79 (-0.85, -0.73) | 7.81 (6.10) | 7.87 (5.89) | -0.06 (-0.15, 0.03) |
| median [IQR] | 6.00 [4.00, 10.00] | 7.00 [4.00, 11.00] | - (-, -) | 6.00 [4.00, 10.00] | 6.00 [4.00, 10.00] | - (-, -) |
| min, max | 0.00, 185.00 | 0.00, 107.00 | - (-, -) | 0.00, 94.00 | 0.00, 84.00 | - (-, -) |
| Number of endocrinologist visits | 0.00,100.00 | 0.00,107.00 | (, , | 0.00,01.00 | 0.00,01.00 | ( ) / |
| mean (sd) | 0.26 (1.08) | 0.43 (1.26) | -0.17 (-0.19, -0.16) | 0.34 (1.31) | 0.36 (1.02) | -0.03 (-0.04, -0.01) |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) |
| min, max | 0.00 [0.00, 0.00] | 0.00, 46.00 | - (-, -)<br>- (-, -) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -)<br>- (-, -) |
| | 0.00, 31.00 | 0.00, 40.00 | - (-, -) | 0.00, 31.00 | 0.00, 33.00 | - (-, -) |
| Number of cardiologist visitsmean (sd) | 0.96 (2.68) | 0.90 (2.53) | 0.06 (0.03, 0.09) | 0.88 (2.41) | 0.91 (2.52) | -0.04 (-0.07, 0.00) |
| mean (sd)median [IQR] | 0.96 (2.68) | 0.90 (2.53) | - (-, -) | 0.88 (2.41) | 0.91 (2.52) | |
| | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | - (-, -)<br>- (-, -) | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | - (-, -)<br>- (-, -) |
| min, max | 0.00, 97.00 | 0.00, 136.00 | - (-, -) | 0.00, 70.00 | 0.00, 85.00 | - (-, -) |
| Number of internal/family medicine visits | 5.07 (0.00) | 1.00 (5.00) | 0.55 (0.40.004) | 500 (550) | 5.00 (5.00) | 0.00/.040.000 |
| mean (sd) | 5.37 (6.38) | 4.82 (5.29) | 0.55 (0.49, 0.61) | 5.00 (5.56) | 5.08 (5.60) | -0.08 (-0.16, 0.01) |
| median [IQR] | 4.00 [2.00, 7.00] | 4.00 [2.00, 6.00] | - (-, -) | 4.00 [2.00, 6.00] | 4.00 [2.00, 7.00] | - (-, -) |
| min, max | 0.00, 159.00 | 0.00, 178.00 | - (-, -) | 0.00, 121.00 | 0.00, 120.00 | - (-, -) |
| Number of Electrocardiograms (ECG/EKG) | | | | | | |
| mean (sd) | 0.81 (1.65) | 0.72 (1.35) | 0.09 (0.07, 0.10) | 0.74 (1.37) | 0.75 (1.40) | -0.01 (-0.03, 0.01) |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | - (-, -) | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | - (-, -) |
| min, max | 0.00, 173.00 | 0.00, 35.00 | - (-, -) | 0.00, 31.00 | 0.00, 35.00 | - (-, -) |
| Number of Echocardiograms | | | | | | |
| mean (sd) | 0.23 (0.65) | 0.21 (0.62) | 0.02 (0.01, 0.02) | 0.21 (0.59) | 0.21 (0.60) | -0.01 (-0.02, 0.00) |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) |
| min, max | 0.00, 13.00 | 0.00, 22.00 | - (-, -) | 0.00, 13.00 | 0.00, 11.00 | - (-, -) |
| Out-of-pocket medication cost | | | | | | |
| mean (sd) | 389.99 (559.90) | 480.98 (813.50) | -90.99 (-97.66, -84.32) | 429.65 (662.77) | 434.85 (595.56) | -5.20 (-14.79, 4.39) |
| median [IQR] | 253.61 [105.46, 500.00] | 285.52 [110.00, 611.65] | - (-, -) | 266.10 [106.07, 551.39] | 271.43 [110.00, 573.55] | - (-, -) |
| min, max | -8,410.21, 33,692.27 | -26,088.85, 62,075.17 | - (-, -) | -8,410.21, 33,692.27 | -19,471.05, 19,642.72 | - (-, -) |
| Unique brand medicines | | | | | | |
| mean (sd) | 12.20 (6.21) | 13.44 (6.62) | -1.24 (-1.31, -1.18) | 12.64 (6.51) | 12.70 (6.07) | -0.06 (-0.15, 0.04) |
| median [IQR] | 11.00 [8.00, 15.00] | 12.00 [9.00, 17.00] | - (-, -) | 11.00 [8.00, 16.00] | 12.00 [8.00, 16.00] | - (-, -) |
| min, max | 1.00, 69,00 | 1.00, 74.00 | - (-, -) | 1.00, 69,00 | 1.00, 63.00 | - (-, -) |
| Unique generic medicines | | | · · · · | | | ( ) / |
| mean (sd) | 11.96 (6.02) | 13.17 (6.44) | -1.21 (-1.27, -1.15) | 12.39 (6.31) | 12.46 (5.91) | -0.07 (-0.16, 0.03) |
| median [IQR] | 11.00 [8.00, 15.00] | 12.00 [9.00, 17.00] | - (-, -) | 11.00 [8.00, 16.00] | 11.00 [8.00, 16.00] | - (-, -) |
| min, max | 1.00, 66.00 | 1.00, 72.00 | - (-, -) | 1.00, 66.00 | 1.00, 62.00 | - (-, -)<br>- (-, -) |
| Colonoscopy Sigmoidoscopy; n (%) | 2.00,00.00 | | | | | 111 |
| | 5.892 (9.4%) | 10.417 (10.3%) | -0.9% (-1.2% -0.6%) | 3 195 (9 6%) | 3 207 (9 7%) | -0.0% (-0.5% 0.4%) |
| | 5,892 (9.4%) | 10,417 (10.3%) | -0.9% (-1.2%, -0.6%) | 3,195 (9.6%) | 3,207 (9.7%) | -0.0% (-0.5%, 0.4%) |
| Flu Pneumococcal vaccine; n (%) | 19,898 (31.9%) | 29,026 (28.8%) | 3.1% (2.6%, 3.5%) | 10,109 (30.5%) | 10,040 (30.3%) | 0.2% (-0.5%, 0.9%) |
| Pap smear; n (%) | 19,898 (31.9%)<br>5,815 (9.3%) | 29,026 (28.8%)<br>12,717 (12.6%) | 3.1% (2.6%, 3.5%)<br>-3.3% (-3.6%, -3.0%) | 10,109 (30.5%)<br>3,589 (10.8%) | 10,040 (30.3%)<br>3,596 (10.8%) | 0.2% (-0.5%, 0.9%)<br>-0.0% (-0.5%, 0.5%) |
| Pap smear, n (%) PSA test, n (%) | 19,898 (31.9%)<br>5,815 (9.3%)<br>13,757 (22.0%) | 29,026 (28.8%)<br>12,717 (12.6%)<br>19,787 (19.6%) | 3.1% (2.6%, 3.5%)<br>-3.3% (-3.6%, -3.0%)<br>2.4% (2.0%, 2.8%) | 10,109 (30.5%)<br>3,589 (10.8%)<br>7,069 (21.3%) | 10,040 (30.3%)<br>3,596 (10.8%)<br>7,046 (21.2%) | 0.2% (-0.5%, 0.9%)<br>-0.0% (-0.5%, 0.5%)<br>0.1% (-0.6%, 0.7%) |
| Pap smear, n (%) PSA test; n (%) Fecal occult blood test; n (%) | 19,898 (31.9%)<br>5,815 (9.3%)<br>13,757 (22.0%)<br>3,407 (5.5%) | 29,026 (28.8%)<br>12,717 (12.6%)<br>19,787 (19.6%)<br>3,797 (3.8%) | 3.1% (2.6%, 3.5%)<br>-3.3% (-3.6%, -3.0%)<br>2.4% (2.0%, 2.8%)<br>1.7% (1.5%, 1.9%) | 10,109 (30.5%)<br>3,589 (10.8%)<br>7,069 (21.3%)<br>1,520 (4.6%) | 10,040 (30.3%)<br>3,596 (10.8%)<br>7,046 (21.2%)<br>1,518 (4.6%) | 0.2% (-0.5%, 0.9%)<br>-0.0% (-0.5%, 0.5%)<br>0.1% (-0.6%, 0.7%)<br>0.0% (-0.3%, 0.3%) |
| Pap smear, n (%) PSA test n (%) Fecal occult blood test n (%) Bone mineral density tests; n (%) | 19,898 (31.9%)<br>5,815 (9.3%)<br>13,757 (22.0%)<br>3,407 (5.5%)<br>1,940 (3.1%) | 29,026 (28.8%)<br>12,717 (12.6%)<br>19,787 (19.6%)<br>3,797 (3.8%)<br>3,229 (3.2%) | 3.1% (2.6%, 3.5%)<br>-3.3% (-3.6%, -3.0%)<br>2.4% (2.0%, 2.8%)<br>1.7% (1.5%, 1.9%)<br>-0.1% (-0.3%, 0.1%) | 10,109 (30.5%)<br>3,589 (10.8%)<br>7,069 (21.3%)<br>1,520 (4.6%)<br>1,055 (3.2%) | 10,040 (30.3%)<br>3,596 (10.8%)<br>7,046 (21.2%)<br>1,518 (4.6%)<br>1,038 (3.1%) | 0.2% (-0.5%, 0.9%)<br>-0.0% (-0.5%, 0.5%)<br>0.1% (-0.6%, 0.7%)<br>0.0% (-0.3%, 0.3%)<br>0.1% (-0.2%, 0.3%) |
| Pap smear, n (%) PSA test n (%) Feal occult blood test, n (%) Bone mineral density tests; n (%) Mammograms; n (%) | 19,898 (31.9%)<br>5,815 (9.3%)<br>13,757 (22.0%)<br>3,407 (5.5%)<br>1,940 (3.1%)<br>12,630 (20.2%) | 29,026 (28.8%)<br>12,717 (12.6%)<br>19,787 (19.6%)<br>3,797 (3.8%)<br>3,229 (3.2%)<br>26,469 (26.2%) | 3.1% (2.6%, 3.5%)<br>3.3% (3.6%, 3.0%)<br>2.4% (2.0%, 2.8%)<br>1.7% (1.5%, 1.9%)<br>-0.1% (-0.3%, 0.1%)<br>-6.0% (-6.4%, -5.6%) | 10,109 (30.5%)<br>3,589 (10.8%)<br>7,069 (21.3%)<br>1,520 (4.6%)<br>1,055 (3.2%)<br>7,642 (23.0%) | 10,040 (30,3%)<br>3,596 (10,8%)<br>7,046 (21,2%)<br>1,518 (4,6%)<br>1,038 (31%)<br>7,624 (23,0%) | 0.2% (-0.5%, 0.9%)<br>-0.0% (-0.5%, 0.5%)<br>0.1% (-0.6%, 0.7%)<br>0.0% (-0.3%, 0.3%)<br>0.1% (-0.2%, 0.3%)<br>0.1% (-0.6%, 0.7%) |
| Pap smear, n (%) PSA test; n (%) Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) | 19,898 (31.9%)<br>5,815 (9.3%)<br>13,757 (22.0%)<br>3,407 (5.5%)<br>1,940 (3.1%) | 29,026 (28.8%)<br>12,717 (12.6%)<br>19,787 (19.6%)<br>3,797 (3.8%)<br>3,229 (3.2%) | 3.1% (2.6%, 3.5%)<br>-3.3% (-3.6%, -3.0%)<br>2.4% (2.0%, 2.8%)<br>1.7% (1.5%, 1.9%)<br>-0.1% (-0.3%, 0.1%) | 10,109 (30.5%)<br>3,589 (10.8%)<br>7,069 (21.3%)<br>1,520 (4.6%)<br>1,055 (3.2%) | 10,040 (30.3%)<br>3,596 (10.8%)<br>7,046 (21.2%)<br>1,518 (4.6%)<br>1,038 (3.1%) | 0.2% (-0.5%, 0.9%)<br>-0.0% (-0.5%, 0.5%)<br>0.1% (-0.6%, 0.7%)<br>0.0% (-0.3%, 0.3%)<br>0.1% (-0.2%, 0.3%) |
| Pap smear, n (%) PSA test; n (%) Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbAIC tests | 19,898 (31.9%) 5,815 (9.3%) 13,757 (22.0%) 3,407 (5.5%) 1,940 (3.1%) 12,630 (20.2%) 9,901 (15.9%) | 29,026 (28.8%)<br>12,717 (12.6%)<br>19,787 (19.6%)<br>3,797 (3.8%)<br>3,229 (3.2%)<br>26,469 (26.2%)<br>32,017 (31.7%) | 3.1% (2.6%, 3.5%) -3.3% (-3.6%, -3.0%) 2.4% (2.0%, 2.8%) 1.7% (1.5%, 1.9%) -0.1% (-0.3%, 0.1%) -6.0% (-6.4%, -5.6%) -15.9% (-16.3%, -15.5%) | 10,109 (30.5%)<br>3,589 (10.8%)<br>7,069 (21.3%)<br>1,520 (4.6%)<br>1,055 (3.2%)<br>7,642 (23.0%)<br>7,916 (23.9%) | 10,040 (30.3%)<br>3.596 (10.8%)<br>7,046 (21.2%)<br>1.518 (4.6%)<br>1,038 (3.1%)<br>7,624 (23.0%)<br>7,900 (23.8%) | 0.2% (-0.5%, 0.9%)<br>-0.0% (-0.5%, 0.5%)<br>-0.1% (-0.6%, 0.7%)<br>-0.0% (-0.3%, 0.3%)<br>-0.1% (-0.2%, 0.3%)<br>-0.1% (-0.6%, 0.7%)<br>-0.0% (-0.6%, 0.7%) |
| Pap smear, n (%) PSA test; n (%) Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbA1C testsmean (sd) | 19,898 (31.9%) 5,815 (9.3%) 13,757 (22.0%) 3,407 (5.5%) 1,940 (3.1%) 12,630 (20.2%) 9,901 (15.9%) | 29,026 (28.8%) 12,717 (12.6%) 19,787 (19.6%) 3,797 (3.8%) 3,229 (3.2%) 26,469 (26.2%) 32,017 (31.7%) | 3.1% (2.6%, 3.5%) -3.3% (-3.6%, -3.0%) 2.4% (2.0%, 2.8%) 1.7% (1.5%, 1.9%) -0.1% (-0.3%, 0.1%) -6.0% (-6.4%, -5.6%) -15.9% (-16.3%, -15.5%) | 10,109 (30.5%)<br>3,589 (10.8%)<br>7,069 (21.3%)<br>1,520 (4.6%)<br>1,055 (3.2%)<br>7,642 (23.0%)<br>7,916 (23.9%) | 10,040 (30,3%) 3,596 (10,8%) 7,046 (21,2%) 1,518 (4,6%) 1,038 (3,1%) 7,624 (23,0%) 7,900 (23,8%) | 0.2% (-0.5%, 0.9%) -0.0% (-0.5%, 0.5%) 0.1% (-0.6%, 0.7%) 0.0% (-0.3%, 0.3%) 0.1% (-0.6%, 0.7%) 0.1% (-0.6%, 0.7%) 0.0% (-0.6%, 0.7%) -0.0( (-0.6%, 0.7%) |
| Pap smear; n (%) PSA test: n (%) Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbAIC testsmean (sd)median [IQR] | 19,898 (31.9%) 5,815 (9.3%) 13,757 (22.0%) 3,407 (5.5%) 1,940 (3.1%) 12,630 (20.2%) 9,901 (15.9%) 2.08 (1.54) 2.00 [1.00, 3.00] | 29,026 (28.8%) 12,717 (12.6%) 19,787 (19.6%) 3,797 (3.8%) 3,229 (3.2%) 26,469 (26.2%) 32,017 (31.7%) 2.15 (1.47) 2.00 [1.00, 3.00] | 3.1% (2.6%, 3.5%) -3.3% (-3.6%, -3.0%) 2.4% (2.0%, 2.8%) 1.7% (1.5%, 1.9%) -0.1% (-0.3%, 0.1%) -6.0% (-6.4%, -5.6%) -15.9% (-16.3%, -15.5%) -0.07 (-0.08, -0.05) -(-, -) | 10,109 (30.5%)<br>3,589 (10.8%)<br>7,069 (21.3%)<br>1,520 (4.6%)<br>1,055 (3.2%)<br>7,642 (23.0%)<br>7,916 (23.9%)<br>216 (1.42)<br>2.00 [1.00, 3.00] | 10,040 (30,3%) 3,596 (10,8%) 7,046 (21,2%) 1,518 (4,6%) 1,038 (3,1%) 7,624 (23,0%) 7,900 (23,8%) 2,16 (1,42) 2,00 [1,00,3,00] | 0.2% (-0.5%, 0.9%) -0.0% (-0.5%, 0.5%) 0.1% (-0.6%, 0.7%) 0.0% (-0.3%, 0.3%) 0.1% (-0.2%, 0.3%) 0.1% (-0.6%, 0.7%) 0.0% (-0.6%, 0.7%) -0.01 (-0.6%, 0.02) -(-,-) |
| Pap smear, n (%) PSA test: n (%) Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbAIC testsmean (sd)median [IQR]min, max | 19,898 (31.9%) 5,815 (9.3%) 13,757 (22.0%) 3,407 (5.5%) 1,940 (3.1%) 12,630 (20.2%) 9,901 (15.9%) | 29,026 (28.8%) 12,717 (12.6%) 19,787 (19.6%) 3,797 (3.8%) 3,229 (3.2%) 26,469 (26.2%) 32,017 (31.7%) | 3.1% (2.6%, 3.5%) -3.3% (-3.6%, -3.0%) 2.4% (2.0%, 2.8%) 1.7% (1.5%, 1.9%) -0.1% (-0.3%, 0.1%) -6.0% (-6.4%, -5.6%) -15.9% (-16.3%, -15.5%) | 10,109 (30.5%)<br>3,589 (10.8%)<br>7,069 (21.3%)<br>1,520 (4.6%)<br>1,055 (3.2%)<br>7,642 (23.0%)<br>7,916 (23.9%) | 10,040 (30,3%) 3,596 (10,8%) 7,046 (21,2%) 1,518 (4,6%) 1,038 (3,1%) 7,624 (23,0%) 7,900 (23,8%) | 0.2% (-0.5%, 0.9%) -0.0% (-0.5%, 0.5%) 0.1% (-0.6%, 0.7%) 0.0% (-0.3%, 0.3%) 0.1% (-0.6%, 0.7%) 0.1% (-0.6%, 0.7%) 0.0% (-0.6%, 0.7%) -0.0( (-0.6%, 0.7%) |
| Pap smear; n (%) PSA test: n (%) Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbAIC testsmean (sd)median [IQR] | 19,898 (31.9%) 5,815 (9.3%) 13,757 (22.0%) 3,407 (5.5%) 1,940 (3.1%) 12,630 (20.2%) 9,901 (15.9%) 2.08 (1.54) 2.00 (1.00, 3.00) 0.00, 122.00 | 29,026 (28.8%) 12,717 (12.6%) 19,787 (19.6%) 3,797 (3.8%) 3,229 (3.2%) 26,469 (26.2%) 32,017 (31.7%) 2.15 (1.47) 2.00 [1.00, 3.00] 0.00,151.00 | 3.1% (2.6%, 3.5%) -3.3% (-3.6%, -3.0%) 2.4% (2.0%, 2.8%) 1.7% (1.5%, 1.9%) -0.1% (-0.3%, 0.1%) -6.0% (-6.4%, -5.6%) -15.9% (-16.3%, -15.5%) -0.07 (-0.08, -0.05) -(-, -) -(-, -) | 10,109 (30.5%) 3,589 (10.8%) 7,069 (21.3%) 1,520 (4.6%) 1,055 (3.2%) 7,542 (23.0%) 7,916 (23.9%) 2,16 (1.42) 2,00 (1.00, 3.00) 0,00, 48.00 | 10,040 (30.3%) 3,596 (10.8%) 7,046 (21.2%) 1,518 (4.6%) 1,038 (3.1%) 7,624 (23.0%) 7,900 (23.8%) 2,16 (1.42) 2,00 [1.00, 3.00] 0,00,40.00 | 0.2% (-0.5%, 0.9%) -0.0% (-0.5%, 0.5%) 0.1% (-0.6%, 0.7%) 0.0% (-0.3%, 0.3%) 0.1% (-0.6%, 0.7%) 0.1% (-0.6%, 0.7%) 0.0% (-0.6%, 0.7%) -0.0% (-0.6%, 0.7%) |
| Pap smear, n (%) PSA test: n (%) Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbAIC testsmean (sd)median [IQR]min, max | 19,898 (31.9%) 5,815 (9.3%) 13,757 (22.0%) 3,407 (5.5%) 1,940 (3.1%) 12,630 (20.2%) 9,901 (15.9%) 2.08 (1.54) 2.00 [1.00, 3.00] | 29,026 (28.8%) 12,717 (12.6%) 19,787 (19.6%) 3,797 (3.8%) 3,229 (3.2%) 26,469 (26.2%) 32,017 (31.7%) 2.15 (1.47) 2.00 [1.00, 3.00] | 3.1% (2.6%, 3.5%) -3.3% (-3.6%, -3.0%) 2.4% (2.0%, 2.8%) 1.7% (1.5%, 1.9%) -0.1% (-0.3%, 0.1%) -6.0% (-6.4%, -5.6%) -15.9% (-16.3%, -15.5%) -0.07 (-0.08, -0.05) -(-, -) | 10,109 (30.5%)<br>3,589 (10.8%)<br>7,069 (21.3%)<br>1,520 (4.6%)<br>1,055 (3.2%)<br>7,642 (23.0%)<br>7,916 (23.9%)<br>216 (1.42)<br>2.00 [1.00, 3.00] | 10,040 (30,3%) 3,596 (10,8%) 7,046 (21,2%) 1,518 (4,6%) 1,038 (3,1%) 7,624 (23,0%) 7,900 (23,8%) 2,16 (1,42) 2,00 [1,00,3,00] | 0.2% (-0.5%, 0.9%) -0.0% (-0.5%, 0.5%) 0.1% (-0.6%, 0.7%) 0.0% (-0.3%, 0.3%) 0.1% (-0.2%, 0.3%) 0.1% (-0.6%, 0.7%) 0.0% (-0.6%, 0.7%) -0.01 (-0.6%, 0.02) -(-,-) |
| Pap smear, n (%) PSA test; n (%) Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbA1C testsmean (sd)median [IQR]min, max Lipid panels | 19,898 (31.9%) 5,815 (9.3%) 13,757 (22.0%) 3,407 (5.5%) 1,940 (3.1%) 12,630 (20.2%) 9,901 (15.9%) 2.08 (1.54) 2.00 (1.00, 3.00) 0.00, 122.00 | 29,026 (28.8%) 12,717 (12.6%) 19,787 (19.6%) 3,797 (3.8%) 3,229 (3.2%) 26,469 (26.2%) 32,017 (31.7%) 2.15 (1.47) 2.00 [1.00, 3.00] 0.00,151.00 | 3.1% (2.6%, 3.5%) -3.3% (-3.6%, -3.0%) 2.4% (2.0%, 2.8%) 1.7% (1.5%, 1.9%) -0.1% (-0.3%, 0.1%) -6.0% (-6.4%, -5.6%) -15.9% (-16.3%, -15.5%) -0.07 (-0.08, -0.05) -(-, -) -(-, -) | 10,109 (30.5%) 3,589 (10.8%) 7,069 (21.3%) 1,520 (4.6%) 1,055 (3.2%) 7,542 (23.0%) 7,916 (23.9%) 2,16 (1.42) 2,00 (1.00, 3.00) 0,00, 48.00 | 10,040 (30.3%) 3,596 (10.8%) 7,046 (21.2%) 1,518 (4.6%) 1,038 (3.1%) 7,624 (23.0%) 7,900 (23.8%) 2,16 (1.42) 2,00 [1.00, 3.00] 0,00,40.00 | 0.2% (-0.5%, 0.9%) -0.0% (-0.5%, 0.5%) 0.1% (-0.6%, 0.7%) 0.0% (-0.3%, 0.3%) 0.1% (-0.6%, 0.7%) 0.1% (-0.6%, 0.7%) 0.0% (-0.6%, 0.7%) -0.0% (-0.6%, 0.7%) |
| Pap smear, n (%) PSA test; n (%) FSA test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbA1C testsmean (sd)median [IQR]min, max Upid panelsmean (sd) | 19,898 (31.9%) 5,815 (9.3%) 13,757 (22.0%) 3,407 (5.5%) 1,940 (3.1%) 12,630 (20.2%) 9,901 (15.9%) 2.08 (1.54) 2.00 (1.00, 3.00) 0.00, 122.00 | 29,026 (28.8%) 12,717 (12.6%) 19,787 (19.6%) 3,797 (3.8%) 3,229 (3.2%) 26,469 (26.2%) 32,017 (31.7%) 2.15 (1.47) 2.00 [1.00, 3.00] 0.00,151.00 | 3.1% (2.6%, 3.5%) -3.3% (-3.6%, -3.0%) 2.4% (2.0%, 2.8%) 1.7% (1.5%, 1.9%) -0.1% (-0.3%, 0.1%) -6.0% (-6.4%, -5.6%) -15.9% (-16.3%, -15.5%) -0.07 (-0.08, -0.05) -(-, -) -(-, -) | 10,109 (30.5%) 3,589 (10.8%) 7,069 (21.3%) 1,520 (4.6%) 1,055 (3.2%) 7,642 (23.0%) 7,916 (23.9%) 216 (1.42) 2.00 [1.00, 3.00] 0.00, 48.00 | 10,040 (30,3%) 3,596 (10,8%) 7,046 (21,2%) 1,518 (4,6%) 1,038 (3,1%) 7,624 (23,0%) 7,900 (23,8%) 2.16 (1,42) 2.00 [1,00,3,00] 0.00, 40,00 | 0.2% (-0.5%, 0.9%) -0.0% (-0.5%, 0.5%) 0.1% (-0.6%, 0.7%) 0.1% (-0.6%, 0.7%) 0.0% (-0.3%, 0.3%) 0.1% (-0.6%, 0.7%) 0.0% (-0.6%, 0.7%) -0.01 (-0.0%, 0.02) -(-, -) -(-, -) |
| Pap smear; n (%) PSA test; n (%) Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbA1C testsmean (sd)median [IQR]min, max Lipid panelsmean (sd)median [IQR] | 19,898 (31.9%) 5,815 (9.3%) 13,757 (22.0%) 3,407 (5.5%) 1,940 (3.1%) 12,630 (20.2%) 9,901 (15.9%) 2.08 (1.54) 2.00 [1.00, 3.00] 0.00, 122.00 1.50 (1.36) 1.00 [1.00, 2.00] | 29,026 (28.8%) 12,717 (12.6%) 19,787 (19.6%) 3,797 (3.8%) 3,229 (3.2%) 26,469 (26.2%) 32,017 (31.7%) 2.15 (1.47) 2.00 [1.00, 3.00] 0.00, 151.00 1.55 (1.29) 1.00 [1.00, 2.00] | 3.1% (2.6%, 3.5%) -3.3% (-3.6%, -3.0%) 2.4% (2.0%, 2.8%) 1.7% (1.5%, 1.9%) -0.1% (-0.3%, 0.1%) -6.0% (-6.4%, -5.6%) -15.9% (-16.3%, -15.5%) -0.07 (-0.08, -0.05) -(-, -) -(-, -) -(-, -) | 10,109 (30.5%) 3,589 (10.8%) 7,069 (21.3%) 1,520 (4.6%) 1,055 (3.2%) 7,642 (23.0%) 7,916 (23.9%) 216 (1.42) 2.00 [1.00, 3.00] 0.00, 48.00 1.55 (1.23) 1.00 [1.00, 2.00] | 10,040 (30,3%) 3,596 (10,8%) 7,046 (21,2%) 1,518 (4,6%) 1,038 (3,1%) 7,624 (23,0%) 7,900 (23,8%) 216 (1,42) 2,00 [1,00,3,00] 0,00,40,00 1,55 (1,26) 1,00 [1,00,2,00] | 0.2% (-0.5%, 0.9%) -0.0% (-0.5%, 0.5%) 0.1% (-0.6%, 0.7%) 0.1% (-0.6%, 0.7%) 0.1% (-0.6%, 0.7%) 0.0% (-0.3%, 0.3%) 0.1% (-0.6%, 0.7%) -0.01 (-0.03, 0.02) -(-, -) -(-, -) -(-, -) |
| Pap smear, n (%) PSA test n (%) Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Mammograms; n (%) Telemedicine; n (%) HbA1C testsmean (sd)median [IQR]min, max Lipid panelsmean (sd)median [IQR]median [IQR]median [IQR]median [IQR]median [IQR]median [IQR]median [IQR] | 19,898 (31.9%) 5,815 (9.3%) 13,757 (22.0%) 3,407 (5.5%) 1,940 (3.1%) 12,630 (20.2%) 9,901 (15.9%) 2.08 (1.54) 2.00 (1.00, 3.00) 0.00, 122.00 1.50 (1.36) 1.00 (1.00, 2.00) 0.00, 122.00 | 29,026 (28.8%) 12,717 (12.6%) 19,787 (19.6%) 3,797 (3.8%) 3,229 (3.2%) 26,469 (26.2%) 32,017 (31.7%) 2.15 (1.47) 2.00 [1.00, 3.00] 0.00, 151.00 1.55 (1.29) 1.00 [1.00, 2.00] | 3.1% (2.6%, 3.5%) -3.3% (-3.6%, -3.0%) 2.4% (2.0%, 2.8%) 1.7% (1.5%, 1.9%) -0.1% (-0.3%, 0.1%) -6.0% (-6.4%, -5.6%) -15.9% (-16.3%, -15.5%) -0.07 (-0.08, -0.05) -(-, -) -(-, -) -(-, -) | 10,109 (30.5%) 3,589 (10.8%) 7,069 (21.3%) 1,520 (4.6%) 1,055 (3.2%) 7,642 (23.0%) 7,916 (23.9%) 216 (1.42) 2.00 (1.00, 3.00) 0.00, 48.00 1.55 (1.23) 1.00 (1.00, 2.00) 0.00, 48.00 | 10,040 (30,3%) 3,596 (10,8%) 7,046 (21,2%) 1,518 (4,6%) 1,038 (3,1%) 7,624 (23,0%) 7,900 (23,8%) 216 (1,42) 2.00 [1,00,3,00] 0.00,40,00 1,55 (1,26) 1,00 [1,00,2,00] 0,00,50,00 | 0.2% (-0.5%, 0.9%) -0.0% (-0.5%, 0.5%) 0.1% (-0.6%, 0.7%) 0.1% (-0.6%, 0.7%) 0.1% (-0.6%, 0.7%) 0.0% (-0.3%, 0.3%) 0.1% (-0.6%, 0.7%) -0.01 (-0.03, 0.02) -(-, -) -(-, -) -(-, -) |
| Pap smear, n (%) PSA test: n (%) Fecal occult blood test: n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbALC testsmean (sd)median [lQR]min, max Lipid panelsmean (sd)median [lQR]median [lQR]median [lQR]median [lQR]mean (sd)median [lQR]mein, max Creatinine tests | 19,898 (31.9%) 5,815 (9.3%) 13,757 (22.0%) 3,407 (5.5%) 1,940 (3.1%) 12,630 (20.2%) 9,901 (15.9%) 2.08 (1.54) 2.00 [1.00, 3.00] 0.00, 122.00 1.50 (1.36) 1.00 [1.00, 2.00] | 29,026 (28.8%) 12,717 (12.6%) 19,787 (19.6%) 3,797 (3.8%) 3,229 (3.2%) 26,469 (26.2%) 32,017 (31.7%) 2.15 (1.47) 2.00 [1.00, 3.00] 0.00,151.00 1.55 (1.29) 1.00 [1.00, 2.00] 0.00,149.00 | 3.1% (2.6%, 3.5%) -3.3% (-3.6%, -3.0%) 2.4% (2.0%, 2.8%) 1.7% (1.5%, 1.9%) -0.1% (-0.3%, 0.1%) -6.0% (-6.4%, -5.6%) -15.9% (-16.3%, -15.5%) -0.07 (-0.08, -0.05) -(-, -) -(-, -) -(-, -) -(-, -) -(-, -) -(-, -) | 10,109 (30.5%) 3,589 (10.8%) 7,069 (21.3%) 1,520 (4.6%) 1,055 (3.2%) 7,642 (23.0%) 7,916 (23.9%) 216 (1.42) 2.00 [1.00, 3.00] 0.00, 48.00 1.55 (1.23) 1.00 [1.00, 2.00] | 10,040 (30,3%) 3,596 (10,8%) 7,046 (21,2%) 1,518 (4,6%) 1,038 (3,1%) 7,624 (23,0%) 7,900 (23,8%) 216 (1,42) 2,00 [1,00,3,00] 0,00,40,00 1,55 (1,26) 1,00 [1,00,2,00] | 0.2% (-0.5%, 0.9%) -0.0% (-0.5%, 0.5%) 0.1% (-0.6%, 0.7%) 0.1% (-0.6%, 0.7%) 0.0% (-0.3%, 0.3%) 0.1% (-0.6%, 0.7%) 0.0% (-0.6%, 0.7%) -0.01 (-0.6%, 0.7%) -0.01 (-0.03, 0.02) -(-, -) -(-, -) -(-, -) -(-, -) -(-, -) |

| min, max | 0.00, 19.00 | 0.00, 43.00 | - (-, -) | 0.00, 17.00 | 0.00, 27.00 | - (-, -) |
|---|---|---|---|---|---|---|
| Natriuretic peptide tests | | | | | | |
| mean (sd) | 0.11 (0.95) | 0.12 (0.88) | -0.01 (-0.02, -0.00) | 0.11 (1.01) | 0.11 (0.84) | 0.00 (-0.01, 0.01) |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) |
| min, max | 0.00, 102.00 | 0.00, 90.00 | - (-, -) | 0.00, 102.00 | 0.00, 62.00 | - (-, -) |
| Urine tests | | | | | | |
| mean (sd) | 0.96 (1.77) | 0.90 (1.62) | 0.06 (0.04, 0.07) | 0.94 (1.67) | 0.95 (1.79) | -0.02 (-0.04, 0.01) |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | - (-, -) | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | - (-, -) |
| min, max | 0.00, 86.00 | 0.00, 53.00 | - (-, -) | 0.00, 86.00 | 0.00, 53.00 | - (-, -) |
| Combined comorbidity score | | | | | | |
| mean (sd) | 1.14 (1.93) | 1.00 (1.66) | 0.14 (0.12, 0.15) | 1.02 (1.73) | 1.04 (1.71) | -0.02 (-0.05, 0.01) |
| median [IQR] | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | - (-, -) | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | - (-, -) |
| min, max | -2.00, 17.00 | -2.00, 17.00 | - (-, -) | -2.00, 14.00 | -2.00, 14.00 | - (-, -) |
| Frailty Score | | | | | | |
| mean (sd) | 0.15 (0.05) | 0.14 (0.04) | 0.00 (0.00, 0.00) | 0.14 (0.04) | 0.14 (0.04) | -0.00 (-0.00, 0.00) |
| median [IQR] | 0.14 [0.12, 0.17] | 0.14 [0.12, 0.16] | - (-, -) | 0.13 [0.12, 0.16] | 0.14 [0.12, 0.16] | - (-, -) |
| min, max | 0.03, 0.61 | 0.05, 0.57 | - (-, -) | 0.03, 0.61 | 0.05, 0.57 | - (-, -) |
| Number of Hospitalizations | | | | | | |
| mean (sd) | 6.43 (28.23) | 4.93 (26.63) | 1.50 (1.23, 1.78) | 5.36 (26.49) | 5.64 (33.72) | -0.28 (-0.74, 0.18) |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) |
| min, max | 0.00, 1,868.00 | 0.00, 3,896.00 | - (-, -) | 0.00, 1,868.00 | 0.00, 3,896.00 | - (-, -) |
| Any hospitalization within prior 91 days; n (%) | 3,211 (5.1%) | 2,965 (2.9%) | 2.2% (2.0%, 2.4%) | 1,245 (3.8%) | 1,319 (4.0%) | -0.2% (-0.5%, 0.1%) |
| Any hospitalization within prior 92-365 days; n (%) | 4,658 (7.5%) | 6,625 (6.6%) | 0.9% (0.6%, 1.1%) | 2,181 (6.6%) | 2,243 (6.8%) | -0.2% (-0.6%, 0.2%) |
| Number of hospitalizations (0, 1, 2 or more) | | | | | | |
| < 1; n (%) | 55,378 (88.7%) | 91,922 (91.1%) | -2.5% (-2.8%, -2.2%) | 30,029 (90.5%) | 29,918 (90.1%) | 0.3% (-0.1%, 0.8%) |
| 1 - <2; n (%) | 538 (0.9%) | 735 (0.7%) | 0.1% (0.0%, 0.2%) | 248 (0.7%) | 267 (0.8%) | -0.1% (-0.2%, 0.1%) |
| >= 2; n (%) | 6,541 (10.5%) | 8,212 (8.1%) | 2.3% (2.0%, 2.6%) | 2,912 (8.8%) | 3,004 (9.1%) | -0.3% (-0.7%, 0.2%) |
| Heart failure hospitalization; n (%) | 1,638 (2.6%) | 1,752 (1.7%) | 0.9% (0.7%, 1.0%) | 593 (1.8%) | 665 (2.0%) | -0.2% (-0.4%, -0.0%) |
| ED visit; n (%) | 18,928 (30.3%) | 29,567 (29.3%) | 1.0% (0.5%, 1.5%) | 9,700 (29.2%) | 9,775 (29.5%) | -0.2% (-0.9%, 0.5%) |
| Acute MI; n (%) | 647 (1.0%) | 892 (0.9%) | 0.2% (0.1%, 0.3%) | 287 (0.9%) | 310 (0.9%) | -0.1% (-0.2%, 0.1%) |
| Old MI; n (%) | 1,019 (1.6%) | 1,506 (1.5%) | 0.1% (0.0%, 0.3%) | 479 (1.4%) | 512 (1.5%) | -0.1% (-0.3%, 0.1%) |
| Heart failure; n (%) | 3,892 (6.2%) | 5,305 (5.3%) | 1.0% (0.7%, 1.2%) | 1,724 (5.2%) | 1,789 (5.4%) | -0.2% (-0.5%, 0.1%) |
| Acute heart failure; n (%) | 1,167 (1.9%) | 1,321 (1.3%) | 0.6% (0.4%, 0.7%) | 433 (1.3%) | 480 (1.4%) | -0.1% (-0.3%, 0.0%) |
| Microalbuminuria or proteinuria; n (%) | 2,086 (3.3%) | 3,523 (3.5%) | -0.2% (-0.3%, 0.0%) | 1,125 (3.4%) | 1,170 (3.5%) | -0.1% (-0.4%, 0.1%) |
| Ratio of brand to generic medications | | | | | | |
| mean (sd) | 1.02 (0.05) | 1.02 (0.05) | -0.00 (-0.00, -0.00) | 1.02 (0.05) | 1.02 (0.04) | 0.00 (-0.00, 0.00) |
| median [IQR] | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | - (-, -) | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | - (-, -) |
| min, max | 0.80, 1.75 | 0.80, 2.00 | - (-, -) | 0.83, 1.75 | 0.80, 2.00 | - (-, -) |

Appendix 7. Balance Assessment - Table 1

| MEDICARE | I | | | | | |
|---|---|---|---|---|---|---|
| Variable | Reference: Sitagliptin | Exposure: Semaglutide injection | Difference | Reference: Sitagliptin | Exposure: Semaglutide injection | Difference |
| Number of patients | 63,191 | 14,635 | - () | 12,339 | 12,339 | - () |
| Year of Cohort Entry Date | 00,101 | 11,000 | ( , , | 12,000 | 12,000 | (, , |
| 2018; n (%) | 24,236 (38.4%) | 1,056 (7.2%) | 31.1% (30.6%, 31.7%) | 1,103 (8.9%) | 1,052 (8.5%) | 0.4% (-0.3%, 1.1%) |
| 2019; n (%) | 22,383 (35.4%) | 5,831 (39.8%) | -4.4% (-5.3%, -3.5%) | 5,177 (42.0%) | 5,189 (42.1%) | -0.1% (-1.3%, 1.1%) |
| 2020; n (%) | 16,572 (26.2%) | 7,748 (52.9%) | -26.7% (-27.6%, -25.8%) | 6,059 (49.1%) | 6,098 (49.4%) | -0.3% (-1.6%, 0.9%) |
| Age | | | | | | |
| mean (sd) | 73.98 (6.31) | 71.51 (4.76) | 2.46 (2.37, 2.55) | 71.74 (5.08) | 71.79 (4.88) | -0.05 (-0.17, 0.08) |
| median [IQR] | 73.00 [69.00, 78.00] | 71.00 [68.00, 74.00] | - (-, -) | 71.00 [68.00, 75.00] | 71.00 [68.00, 75.00] | - (-, -) |
| min, max | 65.00, 106.00 | 65.00, 98.00 | - (-, -) | 65.00, 97.00 | 65.00, 98.00 | - (-, -) |
| Gender (male); n (%) | 26,463 (41.9%) | 6,772 (46.3%) | -4.4% (-5.3%, -3.5%) | 5,467 (44.3%) | 5,585 (45.3%) | -1.0% (-2.2%, 0.3%) |
| Race (Recategorized) | | | | | | |
| White; n (%) | 48,071 (76.1%) | 12,226 (83.5%) | -7.5% (-8.2%, -6.8%) | 10,186 (82.6%) | 10,201 (82.7%) | -0.1% (-1.1%, 0.8%) |
| Other; n (%) | 4,740 (7.5%) | 623 (4.3%) | 3.2% (2.9%, 3.6%) | 570 (4.6%) | 564 (4.6%) | 0.0% (-0.5%, 0.6%) |
| Black; n (%) | 8,181 (12.9%) | 1,274 (8.7%) | 4.2% (3.7%, 4.8%) | 1,152 (9.3%) | 1,143 (9.3%) | 0.1% (-0.7%, 0.8%) |
| Unknown / Missing; n (%) | 2,199 (3.5%) | 512 (3.5%) | -0.0% (-0.4%, 0.3%) | 431 (3.5%) | 431 (3.5%) | 0.0% (-0.5%, 0.5%) |
| Region / State | | | | | | |
| Northest; n (%) | 12,489 (19.8%) | 2,368 (16.2%) | 3.6% (2.9%, 4.3%) | 2,018 (16.4%) | 2,059 (16.7%) | -0.3% (-1.3%, 0.6%) |
| Midwest / North central; n (%) | 13,550 (21.4%) | 3,539 (24.2%) | -2.7% (-3.5%, -2.0%) | 2,901 (23.5%) | 2,893 (23.4%) | 0.1% (-1.0%, 1.1%) |
| South; n (%) | 27,343 (43.3%) | 6,779 (46.3%) | -3.1% (-3.9%, -2.2%) | 5,759 (46.7%) | 5,672 (46.0%) | 0.7% (-0.5%, 2.0%) |
| West; n (%) | 9,708 (15.4%) | 1,943 (13.3%) | 2.1% (1.5%, 2.7%) | 1,655 (13.4%) | 1,710 (13.9%) | -0.4% (-1.3%, 0.4%) |
| Missing, n (%) | 101 (0.2%) | 6 (0.0%) | 0.1% (0.1%, 0.2%) | 6 (0.0%) | 5 (0.0%) | 0.0% (-0.1%, 0.1%) |
| Smoking / Tobacco use; n (%) Weight | 17,742 (28.1%) | 4,116 (28.1%) | -0.0% (-0.9%, 0.8%) | 3,489 (28.3%) | 3,455 (28.0%) | 0.3% (-0.9%, 1.4%) |
| Underweight; n (%) | 86 (0.1%) | 10 (0.1%) | 0.1% (0.0%, 0.1%) | 9 (0.1%) | 9 (0.1%) | 0.0% (-0.1%, 0.1%) |
| Orider weight; n (%) | 1,012 (1.6%) | 77 (0.5%) | 1.1% (0.9%, 1.2%) | 84 (0.7%) | 73 (0.6%) | 0.1% (-0.1%, 0.3%) |
| Overweight; n (%) | 13,555 (21.5%) | 1.829 (12.5%) | 9.0% (8.3%, 9.6%) | 1.645 (13.3%) | 1,718 (13.9%) | -0.6% (-1.5%, 0.3%) |
| Class 1 Obesity; n (%) | 7,601 (12.0%) | 1,435 (9.8%) | 2.2% (1.7%, 2.8%) | 1,281 (10.4%) | 1,307 (10.6%) | -0.2% (-1.0%, 0.6%) |
| Class 2 Obesity; n (%) | 3,537 (5.6%) | 936 (6.4%) | -0.8% (-1.2%, -0.4%) | 813 (6.6%) | 805 (6.5%) | 0.1% (-0.6%, 0.7%) |
| Class 3 Obesity; n (%) | 12,586 (19.9%) | 4,406 (30.1%) | -10.2% (-11.0%, -9.4%) | 3,484 (28.2%) | 3,418 (27.7%) | 0.5% (-0.6%, 1.7%) |
| Unspecified Obesity; n (%) | 24,814 (39.3%) | 5,942 (40.6%) | -1.3% (-2.2%, -0.4%) | 5,023 (40.7%) | 5,009 (40.6%) | 0.1% (-1.1%, 1.3%) |
| Diabetic retinopathy; n (%) | 6,446 (10.2%) | 1,981 (13.5%) | -3.3% (-3.9%, -2.7%) | 1,532 (12.4%) | 1,534 (12.4%) | -0.0% (-0.8%, 0.8%) |
| Diabetic neuropathy; n (%) | 18,998 (30.1%) | 5,175 (35.4%) | -5.3% (-6.2%, -4.4%) | 4,134 (33.5%) | 4,131 (33.5%) | 0.0% (-1.2%, 1.2%) |
| Diabetic nephropathy; n (%) | 17,187 (27.2%) | 4,269 (29.2%) | -2.0% (-2.8%, -1.2%) | 3,418 (27.7%) | 3,443 (27.9%) | -0.2% (-1.3%, 0.9%) |
| Diabetes with other opthalmic complications; n (%) | 1,808 (2.9%) | 404 (2.8%) | 0.1% (-0.2%, 0.4%) | 331 (2.7%) | 340 (2.8%) | -0.1% (-0.5%, 0.3%) |
| Diabetes with peripheral circulatory disorders; n (%) | 8,178 (12.9%) | 2,108 (14.4%) | -1.5% (-2.1%, -0.8%) | 1,678 (13.6%) | 1,665 (13.5%) | 0.1% (-0.8%, 1.0%) |
| Diabetic foot; n (%) | 2,632 (4.2%) | 567 (3.9%) | 0.3% (-0.1%, 0.6%) | 474 (3.8%) | 476 (3.9%) | -0.0% (-0.5%, 0.5%) |
| Erectile dysfunction; n (%) | 1,046 (1.7%) | 356 (2.4%) | -0.8% (-1.1%, -0.5%) | 292 (2.4%) | 285 (2.3%) | 0.1% (-0.3%, 0.4%) |
| Hypoglycemia; n (%) | 8,382 (13.3%) | 2,201 (15.0%) | -1.8% (-2.4%, -1.1%) | 1,824 (14.8%) | 1,759 (14.3%) | 0.5% (-0.4%, 1.4%) |
| Hyperglycemia / DKA / HONK; n (%) | 30,390 (48.1%) | 8,546 (58.4%) | -10.3% (-11.2%, -9.4%) | 6,827 (55.3%) | 6,843 (55.5%) | -0.1% (-1.4%, 1.1%) |
| Skin infections; n (%) | 8,124 (12.9%) | 1,835 (12.5%) | 0.3% (-0.3%, 0.9%) | 1,558 (12.6%) | 1,499 (12.1%) | 0.5% (-0.4%, 1.3%) |
| Stable angina; n (%) | 3,473 (5.5%) | 993 (6.8%) | -1.3% (-1.7%, -0.8%) | 796 (6.5%) | 786 (6.4%) | 0.1% (-0.5%, 0.7%) |
| Unstable angina; n (%) | 2,847 (4.5%) | 705 (4.8%) | -0.3% (-0.7%, 0.1%) | 569 (4.6%) | 558 (4.5%) | 0.1% (-0.4%, 0.6%) |
| Hypertension; n (%) | 56,887 (90.0%) | 12,999 (88.8%) | 1.2% (0.6%, 1.8%) | 10,965 (88.9%) | 10,953 (88.8%) | 0.1% (-0.7%, 0.9%) |
| Hypotension; n (%) | 3,687 (5.8%) | 683 (4.7%)<br>11,366 (77.7%) | 1.2% (0.8%, 1.6%) | 559 (4.5%)<br>9,522 (77.2%) | 571 (4.6%)<br>9,535 (77.3%) | -0.1% (-0.6%, 0.4%) |
| Hyperlipidemia; n (%) Atrial fibrillation: n (%) | 48,759 (77.2%)<br>12.711 (20.1%) | 2.694 (18.4%) | -0.5% (-1.3%, 0.3%)<br>1.7% (1.0%, 2.4%) | 9,522 (77.2%)<br>2.257 (18.3%) | 9,535 (77.3%)<br>2.250 (18.2%) | -0.1% (-1.2%, 0.9%)<br>0.1% (-0.9%, 1.0%) |
| Cardiac conduction disorder; n (%) | 6,039 (9.6%) | 1,268 (8.7%) | 0.9% (0.4%, 1.4%) | 1,056 (8.6%) | 1,077 (8.7%) | -0.2% (-0.9%, 1.0%) |
| Previous cardiac procedure (CABG, PTCA, Stent); n (%) | 1,994 (3.2%) | 598 (4.1%) | -0.9% (-1.3%, -0.6%) | 468 (3.8%) | 470 (3.8%) | -0.2% (-0.5%, 0.5%) |
| Ischemic stroke; n (%) | 1,900 (3.0%) | 260 (1.8%) | 1.2% (1.0%, 1.5%) | 256 (2.1%) | 232 (1.9%) | 0.2% (-0.2%, 0.6%) |
| PVD diagnosis or surgery; n (%) | 8,676 (13.7%) | 1,883 (12.9%) | 0.9% (0.3%, 1.5%) | 1,551 (12.6%) | 1,558 (12.6%) | -0.1% (-0.9%, 0.8%) |
| Other cardiac dysrhythmia; n (%) | 16,974 (26.9%) | 3,614 (24.7%) | 2.2% (1.4%, 3.0%) | 3,048 (24.7%) | 3,008 (24.4%) | 0.3% (-0.8%, 1.4%) |
| Cardiomyopathy; n (%) | 4,617 (7.3%) | 1,091 (7.5%) | -0.1% (-0.6%, 0.3%) | 859 (7.0%) | 910 (7.4%) | -0.4% (-1.1%, 0.2%) |
| Valve disorders; n (%) | 10,141 (16.0%) | 2,123 (14.5%) | 1.5% (0.9%, 2.2%) | 1,770 (14.3%) | 1,774 (14.4%) | -0.0% (-0.9%, 0.9%) |
| Valve replacement; n (%) | 1,507 (2.4%) | 363 (2.5%) | -0.1% (-0.4%, 0.2%) | 309 (2.5%) | 300 (2.4%) | 0.1% (-0.3%, 0.5%) |
| TIA; n (%) | 2,087 (3.3%) | 340 (2.3%) | 1.0% (0.7%, 1.3%) | 299 (2.4%) | 290 (2.4%) | 0.1% (-0.3%, 0.5%) |
| Edema; n (%) | 10,680 (16.9%) | 2,427 (16.6%) | 0.3% (-0.4%, 1.0%) | 1,998 (16.2%) | 1,979 (16.0%) | 0.2% (-0.8%, 1.1%) |
| Venous thromboembolism / Pulmonary embolism; n (%) | 3,010 (4.8%) | 650 (4.4%) | 0.3% (-0.1%, 0.7%) | 534 (4.3%) | 548 (4.4%) | -0.1% (-0.6%, 0.4%) |
| Pulmonary hypertension; n (%) | 3,165 (5.0%) | 590 (4.0%) | 1.0% (0.6%, 1.3%) | 489 (4.0%) | 498 (4.0%) | -0.1% (-0.6%, 0.4%) |
| Implantable cardioverter defibrillator; n (%) | 390 (0.6%) | 81 (0.6%) | 0.1% (-0.1%, 0.2%) | 66 (0.5%) | 75 (0.6%) | -0.1% (-0.3%, 0.1%) |
| Hyperkalemia; n (%) | 1,349 (2.1%) | 241 (1.6%) | 0.5% (0.2%, 0.7%) | 217 (1.8%) | 210 (1.7%) | 0.1% (-0.3%, 0.4%) |
| Coronary atherosclerosis; n (%) | 22,046 (34.9%) | 5,363 (36.6%) | -1.8% (-2.6%, -0.9%) | 4,307 (34.9%) | 4,357 (35.3%) | -0.4% (-1.6%, 0.8%) |
| Cerebrovascular procedure; n (%) | 265 (0.4%) | 48 (0.3%) | 0.1% (-0.0%, 0.2%) | 56 (0.5%) | 43 (0.3%) | 0.1% (-0.1%, 0.3%) |
| Insertion of pacemakers / removal of cardiac lead; n (%) | 381 (0.6%) | 53 (0.4%) | 0.2% (0.1%, 0.4%) | 49 (0.4%) | 43 (0.3%) | 0.0% (-0.1%, 0.2%) |
|---|---|---|---|---|---|---|
| CKD stage 1-2; n (%) | 2,704 (4.3%) | 628 (4.3%) | -0.0% (-0.4%, 0.4%) | 512 (4.1%) | 516 (4.2%) | -0.0% (-0.5%, 0.5%) |
| CKD stage 3-4; n (%) | 13,570 (21.5%) | 3,364 (23.0%) | -1.5% (-2.3%, -0.8%) | 2,691 (21.8%) | 2,708 (21.9%) | -0.1% (-1.2%, 0.9%) |
| Unspecified CKD; n (%) | 6,892 (10.9%) | 1,466 (10.0%) | 0.9% (0.3%, 1.4%) | 1,196 (9.7%) | 1,204 (9.8%) | -0.1% (-0.8%, 0.7%) |
| Acute kidney injury; n (%) | 9,378 (14.8%) | 1,671 (11.4%) | 3.4% (2.8%, 4.0%) | 1,459 (11.8%) | 1,427 (11.6%) | 0.3% (-0.6%, 1.1%) |
| Hypertensive nephropathy; n (%) | 12.874 (20.4%) | 2.924 (20.0%) | 0.4% (-0.3%, 1.1%) | 2.354 (19.1%) | 2,386 (19.3%) | -0.3% (-1.3%, 0.7%) |
| Urinary tract infections; n (%) | 14,898 (23.6%) | 2,823 (19.3%) | 4.3% (3.6%, 5.0%) | 2,485 (20.1%) | 2,452 (19.9%) | 0.3% (-0.7%, 1.3%) |
| Genital infections; n (%) | 1,930 (3.1%) | 434 (3.0%) | 0.1% (-0.2%, 0.4%) | 369 (3.0%) | 356 (2.9%) | 0.1% (-0.3%, 0.5%) |
| Urolithiasis (Kidney and urinary stone); n (%) | 3.258 (5.2%) | 762 (5.2%) | -0.1% (-0.5%, 0.4%) | 632 (5.1%) | 649 (5.3%) | -0.1% (-0.7%, 0.4%) |
| COPD; n (%) | 12,124 (19.2%) | 2,595 (17.7%) | 1.5% (0.8%, 2.1%) | 2,195 (17.8%) | 2,221 (18.0%) | -0.2% (-1.2%, 0.8%) |
| Asthma; n (%) | 6,824 (10.8%) | 1,622 (11.1%) | -0.3% (-0.9%, 0.3%) | 1,340 (10.9%) | 1,350 (10.9%) | -0.1% (-0.9%, 0.7%) |
| Obstructive sleep apnea; n (%) | 14,082 (22.3%) | 4,895 (33.4%) | -11.2% (-12.0%, -10.3%) | 3,846 (31.2%) | 3,811 (30.9%) | 0.3% (-0.9%, 1.4%) |
| Serious bacterial infections; n (%) | 5,266 (8.3%) | 775 (5.3%) | 3.0% (2.6%, 3.5%) | 710 (5.8%) | 688 (5.6%) | 0.2% (-0.4%, 0.8%) |
| Pneumonia; n (%) | 5,836 (9.2%) | 1,023 (7.0%) | 2.2% (1.8%, 2.7%) | 861 (7.0%) | 880 (7.1%) | -0.2% (-0.8%, 0.5%) |
| Liver disease; n (%) | 6,984 (11.1%) | 1,763 (12.0%) | -1.0% (-1.6%, -0.4%) | 1,419 (11.5%) | 1,426 (11.6%) | -0.1% (-0.9%, 0.7%) |
| MASH/MASLD; n (%) | 3,097 (4.9%) | 938 (6.4%) | -1.5% (-1.9%, -1.1%) | 735 (6.0%) | 746 (6.0%) | -0.1% (-0.7%, 0.5%) |
| Fractures / Falls; n (%) | 3,040 (4.8%) | 572 (3.9%) | 0.9% (0.5%, 1.3%) | 475 (3.8%) | 492 (4.0%) | -0.1% (-0.6%, 0.4%) |
| Osteoporosis; n (%) | 4,553 (7.2%) | 906 (6.2%) | 1.0% (0.6%, 1.5%) | 785 (6.4%) | 785 (6.4%) | 0.0% (-0.6%, 0.6%) |
| Osteoarthritis; n (%) | 22,977 (36.4%) | 5,334 (36.4%) | -0.1% (-1.0%, 0.8%) | 4,426 (35.9%) | 4,491 (36.4%) | -0.5% (-1.7%, 0.7%) |
| Depression; n (%) | 12,721 (20.1%) | 2,995 (20.5%) | -0.3% (-1.1%, 0.4%) | 2,549 (20.7%) | 2,508 (20.3%) | 0.3% (-0.7%, 1.3%) |
| Dementia; n (%) | 6,422 (10.2%) | 741 (5.1%) | 5.1% (4.7%, 5.5%) | 697 (5.6%) | 679 (5.5%) | 0.1% (-0.4%, 0.7%) |
| Delirium or psychosis; n (%) | 1,963 (3.1%) | 246 (1.7%) | 1.4% (1.2%, 1.7%) | 241 (2.0%) | 223 (1.8%) | 0.1% (-0.2%, 0.5%) |
| Anxiety; n (%) | 9,888 (15.6%) | 2,195 (15.0%) | 0.6% (0.0%, 1.3%) | 1,885 (15.3%) | 1,886 (15.3%) | -0.0% (-0.9%, 0.9%) |
| * * * * | | 5.064 (34.6%) | 0.5% (-0.4%, 1.3%) | 4,286 (34.7%) | 4,258 (34.5%) | 0.2% (-1.0%, 1.4%) |
| Sleep disorders; n (%) | 22,151 (35.1%) | 3,645 (24.9%) | 4.5% (3.7%, 5.3%) | | 3,116 (25.3%) | -0.2% (-1.0%, 1.4%) |
| Anemia; n (%) | 18,582 (29.4%) | | | 3,096 (25.1%) | | |
| Influenza; n (%) | 1,699 (2.7%) | 281 (1.9%) | 0.8% (0.5%, 1.0%) | 259 (2.1%) | 254 (2.1%) | 0.0% (-0.3%, 0.4%) |
| COVID; n (%) | 306 (0.5%) | 88 (0.6%) | -0.1% (-0.3%, 0.0%) | 69 (0.6%) | 73 (0.6%) | -0.0% (-0.2%, 0.2%) |
| Hyperthyroidism and other thyroid gland disorders; n (%) | 17,605 (27.9%) | 4,302 (29.4%) | -1.5% (-2.4%, -0.7%) | 3,577 (29.0%) | 3,594 (29.1%) | -0.1% (-1.3%, 1.0%) |
| Hypothyroidism; n (%) | 14,477 (22.9%) | 3,542 (24.2%) | -1.3% (-2.1%, -0.5%) | 2,945 (23.9%) | 2,955 (23.9%) | -0.1% (-1.2%, 1.0%) |
| Nephrotic syndrome; n (%) | 55 (0.1%) | 15 (0.1%) | -0.0% (-0.1%, 0.0%) | 13 (0.1%) | 13 (0.1%) | 0.0% (-0.1%, 0.1%) |
| Urinary incontinence; n (%) | 4,406 (7.0%) | 922 (6.3%) | 0.7% (0.2%, 1.1%) | 801 (6.5%) | 793 (6.4%) | 0.1% (-0.6%, 0.7%) |
| Biliary disease; n (%) | 282 (0.4%) | 39 (0.3%) | 0.2% (0.1%, 0.3%) | 30 (0.2%) | 31 (0.3%) | -0.0% (-0.1%, 0.1%) |
| Pancreatitis; n (%) | 149 (0.2%) | 15 (0.1%) | 0.1% (0.1%, 0.2%) | 12 (0.1%) | 14 (0.1%) | -0.0% (-0.1%, 0.1%) |
| Pancreatitis; n (%) Bowel obstruction; n (%) | 149 (0.2%)<br>167 (0.3%) | 15 (0.1%)<br>36 (0.2%) | 0.1% (0.1%, 0.2%)<br>0.0% (-0.1%, 0.1%) | 12 (0.1%)<br>34 (0.3%) | 14 (0.1%)<br>29 (0.2%) | -0.0% (-0.1%, 0.1%)<br>0.0% (-0.1%, 0.2%) |
| Bowel obstruction; n (%) | 167 (0.3%) | 36 (0.2%) | 0.0% (-0.1%, 0.1%) | 34 (0.3%) | 29 (0.2%) | 0.0% (-0.1%, 0.2%) |
| Bowel obstruction; n (%) Gastroparesis; n (%) | | | | | | |
| Bowel obstruction; n (%) Gastroparesis; n (%) Number of antidiabetic drugs on CED | 167 (0.3%)<br>533 (0.8%) | 36 (0.2%)<br>107 (0.7%) | 0.0% (-0.1%, 0.1%)<br>0.1% (-0.0%, 0.3%) | 34 (0.3%)<br>89 (0.7%) | 29 (0.2%)<br>89 (0.7%) | 0.0% (-0.1%, 0.2%)<br>0.0% (-0.2%, 0.2%) |
| Bowel obstruction; n (%) Gastroparesis; n (%) Number of antidiabetic drugs on CEDmean (sd) | 167 (0.3%)<br>533 (0.8%)<br>2.19 (0.83) | 36 (0.2%)<br>107 (0.7%)<br>2.32 (0.90) | 0.0% (-0.1%, 0.1%)<br>0.1% (-0.0%, 0.3%)<br>-0.12 (-0.14, -0.11) | 34 (0.3%)<br>89 (0.7%)<br>2.29 (0.89) | 29 (0.2%)<br>89 (0.7%)<br>2.28 (0.89) | 0.0% (-0.1%, 0.2%)<br>0.0% (-0.2%, 0.2%)<br>0.01 (-0.01, 0.04) |
| Bowel obstruction; n (%) Gastroparesis; n (%) Number of antidiabetic drugs on CEDmean (sd)median [IQR] | 167 (0.3%)<br>533 (0.8%)<br>2.19 (0.83)<br>2.00 [2.00, 3.00] | 36 (0.2%)<br>107 (0.7%)<br>2.32 (0.90)<br>2.00 [2.00, 3.00] | 0.0% (-0.1%, 0.1%)<br>0.1% (-0.0%, 0.3%)<br>-0.12 (-0.14, -0.11)<br>- (-, -) | 34 (0.3%)<br>89 (0.7%)<br>2.29 (0.89)<br>2.00 [2.00, 3.00] | 29 (0.2%)<br>89 (0.7%)<br>2.28 (0.89)<br>2.00 [2.00, 3.00] | 0.0% (-0.1%, 0.2%)<br>0.0% (-0.2%, 0.2%)<br>0.01 (-0.01, 0.04)<br>- (-, -) |
| Bowel obstruction; n (%) Gastroparesis; n (%) Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max | 167 (0.3%)<br>533 (0.8%)<br>2.19 (0.83)<br>2.00 [2.00, 3.00]<br>1.00, 6.00 | 36 (0.2%)<br>107 (0.7%)<br>2.32 (0.90)<br>2.00 (2.00, 3.00)<br>1.00, 6.00 | 0.0% (-0.1%, 0.1%)<br>0.1% (-0.0%, 0.3%)<br>-0.12 (-0.14, -0.11)<br>-(-, -) | 34 (0.3%)<br>89 (0.7%)<br>2.29 (0.89)<br>2.00 [2.00, 3.00]<br>1.00, 6.00 | 29 (0.2%)<br>89 (0.7%)<br>228 (0.89)<br>200 (2.00, 3.00)<br>1.00, 6.00 | 0.0% (-0.1%, 0.2%)<br>0.0% (-0.2%, 0.2%)<br>0.01 (-0.01, 0.04)<br>-(-, -) |
| Bowel obstruction; n (%) Gastroparesis; n (%) Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) | 167 (0.3%)<br>533 (0.8%)<br>219 (0.83)<br>2.00 [2.00, 3.00]<br>1.00, 6.00<br>36,599 (57.9%) | 36 (0.2%)<br>107 (0.7%)<br>2.32 (0.90)<br>2.00 [2.00, 3.00]<br>1.00, 6.00<br>7,195 (49.2%) | 0.0% (-0.1%, 0.1%)<br>0.1% (-0.0%, 0.3%)<br>-0.12 (-0.14, -0.11)<br>-(-, -)<br>-(-, -)<br>8.8% (7.9%, 9.7%) | 34 (0.3%)<br>89 (0.7%)<br>229 (0.89)<br>200 (200, 3.00)<br>1.00, 6.00<br>6,341 (51.4%) | 29 (0.2%)<br>89 (0.7%)<br>228 (0.89)<br>200 (2.00, 3.00)<br>100, 6.00<br>6,364 (51.6%) | 0.0% (-0.1%, 0.2%)<br>0.0% (-0.2%, 0.2%)<br>0.01 (-0.01, 0.04)<br>- (-, -)<br>- (-, -)<br>-0.2% (-1.4%, 1.1%) |
| Bowel obstruction; n (%) Gastroparesis; n (%) Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) | 167 (0.3%)<br>533 (0.8%)<br>219 (0.83)<br>200 [2.00, 3.00]<br>1.00, 6.00<br>36,599 (57.9%)<br>10,558 (16.7%) | 36 (0.2%)<br>107 (0.7%)<br>2.32 (0.90)<br>2.00 (2.00, 3.00)<br>1.00, 6.00<br>7.195 (49.2%)<br>5.854 (40.0%) | 0.0% (-0.1%, 0.1%)<br>0.1% (-0.0%, 0.3%)<br>-0.12 (-0.14, -0.11)<br>-()<br>-()<br>-()<br>-2.3% (-24.1%, -22.4%) | 34 (0.3%)<br>89 (0.7%)<br>2.29 (0.89)<br>2.00 (2.00, 3.00)<br>1.00, 6.00<br>6.341 (51.4%)<br>4.156 (33.7%) | 29 (0.2%)<br>89 (0.7%)<br>2.28 (0.89)<br>2.00 (2.00, 3.00)<br>1.00, 6.00<br>6.364 (51.6%)<br>4,126 (33.4%) | 0.0% (-0.1%, 0.2%)<br>0.0% (-0.2%, 0.2%)<br>0.01 (-0.01, 0.04)<br>-(-,-)<br>-(-,-)<br>-(-,2% (-1.4%, 1.1%)<br>0.2% (-0.9%, 1.4%) |
| Bowel obstruction; n (%) Gastroparesis; n (%) Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) | 167 (0.3%)<br>533 (0.8%)<br>219 (0.83)<br>200 [2.00, 3.00]<br>1.00, 6.00<br>36,599 (57.9%)<br>10,558 [16.7%)<br>20,522 (32.5%) | 36 (0.2%)<br>107 (0.7%)<br>2.32 (0.90)<br>2.00 [2.00, 3.00]<br>1.00, 6.00<br>7,195 (49.2%)<br>5,854 (40.0%)<br>3,386 (23.1%) | 0.0% (-0.1%, 0.1%)<br>0.1% (-0.0%, 0.3%)<br>-0.12 (-0.14, -0.11)<br>-(-,-)<br>-(-,-)<br>8.8% (7.9%, 9.7%)<br>23.3% (-24.1%, -22.4%)<br>9.3% (8.6%, 10.1%) | 34 (0.3%)<br>89 (0.7%)<br>229 (0.89)<br>200 (2.00, 3.00)<br>1.00, 6.00<br>6.341 (51.4%)<br>4.156 (33.7%)<br>3.182 (25.8%) | 29 (0.2%)<br>89 (0.7%)<br>2.28 (0.89)<br>2.00 [2.00, 3.00]<br>1.00, 6.00<br>6.364 (51.6%)<br>4,126 (33.4%)<br>3.097 (25.1%) | 0.0% (-0.1%, 0.2%)<br>0.0% (-0.2%, 0.2%)<br>0.01 (-0.01, 0.04)<br>-(-,-)<br>-(-,-)<br>-0.2% (-1.4%, 1.1%)<br>0.2% (-0.9%, 1.4%)<br>0.7% (-0.4%, 1.8%) |
| Bowel obstruction; n (%) Gastroparesis; n (%) Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of SGLT-2i; n (%) | 167 (0.3%)<br>533 (0.8%)<br>219 (0.83)<br>200 [2.00, 3.00]<br>100, 6.00<br>36,599 (57.9%)<br>10,558 (16.7%)<br>20,522 (32.5%)<br>3,585 (5.7%) | 36 (0.2%)<br>107 (0.7%)<br>2.32 (0.90)<br>2.00 (2.00, 3.00)<br>1.00, 6.00<br>7,195 (49.2%)<br>5,854 (40.0%)<br>3,386 (23.1%)<br>1,880 (12.8%) | 0.0% (-0.1%, 0.1%)<br>0.1% (-0.0%, 0.3%)<br>-0.12 (-0.14, -0.11)<br>-()<br>-()<br>8.8% (7.9%, 9.7%)<br>-23.3% (-24.1%, -22.4%)<br>9.3% (8.6%, 10.1%)<br>-7.2% (-7.7%, -6.6%) | 34 (0.3%)<br>89 (0.7%)<br>229 (0.89)<br>200 (2.00, 3.00)<br>1.00, 6.00<br>6.341 (51.4%)<br>4,156 (33.7%)<br>3,182 (25.5%)<br>1,408 (11.4%) | 29 (0.2%)<br>89 (0.7%)<br>228 (0.89)<br>200 (2.00, 3.00)<br>1.00, 6.00<br>6.364 (51.6%)<br>4,126 (33.4%)<br>3,097 (25.1%)<br>1,361 (11.0%) | 0.0% (-0.1%, 0.2%)<br>0.0% (-0.2%, 0.2%)<br>0.01 (-0.01, 0.04)<br>-(-, -)<br>-(-, -)<br>-(-, -)<br>0.2% (-1.4%, 1.1%)<br>0.2% (-0.9%, 1.4%)<br>0.7% (-0.4%, 1.8%)<br>0.4% (-0.4%, 1.2%) |
| Bowel obstruction; n (%) Gastroparesis; n (%) Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of SGLT-2; n (%) Concomitant use or initiation of SGLT-2; n (%) | 167 (0.3%)<br>533 (0.8%)<br>219 (0.83)<br>200 (2.00, 3.00)<br>1.00, 6.00<br>36,599 (57.9%)<br>10,558 (16.7%)<br>20,522 (32.5%)<br>3,585 (5.7%)<br>4,172 (6.6%) | 36 (0.2%)<br>107 (0.7%)<br>2.32 (0.90)<br>2.00 (2.00, 3.00)<br>1.00, 6.00<br>7.195 (49.2%)<br>5.854 (40.0%)<br>3.386 (23.1%)<br>1.880 (12.8%)<br>975 (6.7%) | 0.0% (-0.1%, 0.1%)<br>0.1% (-0.0%, 0.3%)<br>-0.12 (-0.14, -0.11)<br>-(,-)<br>-(,-)<br>8.8% (7.9%, 9.7%)<br>-23.3% (-24.1%, -22.4%)<br>9.3% (8.6%, 10.1%)<br>-7.2% (-7.7%, -6.6%)<br>-0.1% (-0.5%, 0.4%) | 34 (0.3%)<br>89 (0.7%)<br>229 (0.89)<br>200 (2.00, 3.00)<br>1.00, 6.00<br>6.341 (51.4%)<br>4.156 (33.7%)<br>3.182 (25.8%)<br>1.408 (11.4%)<br>862 (7.0%) | 29 (0.2%)<br>89 (0.7%)<br>228 (0.89)<br>200 (2.00, 3.00)<br>1.00, 6.00<br>6.364 (51.6%)<br>4,126 (33.4%)<br>3,097 (25.1%)<br>1,361 (11.0%)<br>825 (6.7%) | 0.0% (-0.1%, 0.2%)<br>0.0% (-0.2%, 0.2%)<br>0.01 (-0.01, 0.04)<br>-(·, -)<br>-(·, -)<br>-0.2% (-1.4%, 1.1%)<br>0.2% (-0.9%, 1.4%)<br>0.7% (-0.4%, 1.8%)<br>0.4% (-0.4%, 1.2%)<br>0.3% (-0.3%, 0.9%) |
| Bowel obstruction; n (%) Gastroparesis; n (%) Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Past use of Metformin; n (%) | 167 (0.3%)<br>533 (0.8%)<br>219 (0.83)<br>200 [2.00, 3.00]<br>1.00, 6.00<br>36,599 (57.9%)<br>10,558 (16.7%)<br>20,522 (32.5%)<br>3,585 (5.7%)<br>4,172 (6.6%)<br>42,319 (67.0%) | 36 (0.2%)<br>107 (0.7%)<br>2.32 (0.90)<br>2.00 (2.00, 3.00)<br>1.00, 6.00<br>7.195 (49.2%)<br>5.854 (40.0%)<br>3.386 (23.1%)<br>1.880 (12.8%)<br>9.75 (6.7%)<br>9.505 (64.9%) | 0.0% (-0.1%, 0.1%)<br>0.1% (-0.0%, 0.3%)<br>-0.12 (-0.14, -0.11)<br>-(.,-) | 34 (0.3%)<br>89 (0.7%)<br>229 (0.89)<br>200 (2.00, 3.00)<br>1.00, 6.00<br>6.341 (51.4%)<br>4.156 (33.7%)<br>3.182 (25.8%)<br>1,408 (11.4%)<br>862 (7.0%)<br>8,183 (66.3%) | 29 (0.2%)<br>89 (0.7%)<br>2.28 (0.89)<br>2.00 (2.00, 3.00)<br>1.00, 6.00<br>6.364 (51.6%)<br>4.126 (33.4%)<br>3.097 (25.1%)<br>1,361 (11.0%)<br>825 (6.7%)<br>8.174 (66.2%) | 0.0% (-0.1%, 0.2%)<br>0.0% (-0.2%, 0.2%)<br>0.01 (-0.01, 0.04)<br>-(·,·)<br>-(·,·)<br>-(·,·)<br>-(·,·)<br>0.2% (-1.4%, 1.1%)<br>0.2% (-0.9%, 1.4%)<br>0.7% (-0.4%, 1.8%)<br>0.4% (-0.4%, 1.2%)<br>0.3% (-0.3%, 0.9%)<br>0.1% (-1.1%, 1.3%) |
| Bowel obstruction; n (%) Gastroparesis; n (%) Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of SGLT-2; n (%) Concomitant use or initiation of SGLT-2; n (%) | 167 (0.3%)<br>533 (0.8%)<br>219 (0.83)<br>200 (2.00, 3.00)<br>1.00, 6.00<br>36,599 (57.9%)<br>10,558 (16.7%)<br>20,522 (32.5%)<br>3,585 (5.7%)<br>4,172 (6.6%) | 36 (0.2%)<br>107 (0.7%)<br>2.32 (0.90)<br>2.00 (2.00, 3.00)<br>1.00, 6.00<br>7.195 (49.2%)<br>5.854 (40.0%)<br>3.386 (23.1%)<br>1.880 (12.8%)<br>975 (6.7%) | 0.0% (-0.1%, 0.1%)<br>0.1% (-0.0%, 0.3%)<br>-0.12 (-0.14, -0.11)<br>-(,-)<br>-(,-)<br>8.8% (7.9%, 9.7%)<br>-23.3% (-24.1%, -22.4%)<br>9.3% (8.6%, 10.1%)<br>-7.2% (-7.7%, -6.6%)<br>-0.1% (-0.5%, 0.4%) | 34 (0.3%)<br>89 (0.7%)<br>229 (0.89)<br>200 (2.00, 3.00)<br>1.00, 6.00<br>6.341 (51.4%)<br>4.156 (33.7%)<br>3.182 (25.8%)<br>1.408 (11.4%)<br>862 (7.0%) | 29 (0.2%)<br>89 (0.7%)<br>228 (0.89)<br>200 (2.00, 3.00)<br>1.00, 6.00<br>6.364 (51.6%)<br>4,126 (33.4%)<br>3,097 (25.1%)<br>1,361 (11.0%)<br>825 (6.7%) | 0.0% (-0.1%, 0.2%)<br>0.0% (-0.2%, 0.2%)<br>0.01 (-0.01, 0.04)<br>-(·, -)<br>-(·, -)<br>-0.2% (-1.4%, 1.1%)<br>0.2% (-0.9%, 1.4%)<br>0.7% (-0.4%, 1.8%)<br>0.4% (-0.4%, 1.2%)<br>0.3% (-0.3%, 0.9%) |
| Bowel obstruction; n (%) Gastroparesis; n (%) Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Past use of Metformin; n (%) | 167 (0.3%)<br>533 (0.8%)<br>219 (0.83)<br>200 [2.00, 3.00]<br>1.00, 6.00<br>36,599 (57.9%)<br>10,558 (16.7%)<br>20,522 (32.5%)<br>3,585 (5.7%)<br>4,172 (6.6%)<br>42,319 (67.0%) | 36 (0.2%)<br>107 (0.7%)<br>2.32 (0.90)<br>2.00 (2.00, 3.00)<br>1.00, 6.00<br>7.195 (49.2%)<br>5.854 (40.0%)<br>3.386 (23.1%)<br>1.880 (12.8%)<br>9.75 (6.7%)<br>9.505 (64.9%) | 0.0% (-0.1%, 0.1%)<br>0.1% (-0.0%, 0.3%)<br>-0.12 (-0.14, -0.11)<br>-(.,-) | 34 (0.3%)<br>89 (0.7%)<br>229 (0.89)<br>200 (2.00, 3.00)<br>1.00, 6.00<br>6.341 (51.4%)<br>4.156 (33.7%)<br>3.182 (25.8%)<br>1,408 (11.4%)<br>862 (7.0%)<br>8,183 (66.3%) | 29 (0.2%)<br>89 (0.7%)<br>2.28 (0.89)<br>2.00 (2.00, 3.00)<br>1.00, 6.00<br>6.364 (51.6%)<br>4.126 (33.4%)<br>3.097 (25.1%)<br>1,361 (11.0%)<br>825 (6.7%)<br>8.174 (66.2%) | 0.0% (-0.1%, 0.2%)<br>0.0% (-0.2%, 0.2%)<br>0.01 (-0.01, 0.04)<br>-(·,·)<br>-(·,·)<br>-(·,·)<br>-(·,·)<br>0.2% (-1.4%, 1.1%)<br>0.2% (-0.9%, 1.4%)<br>0.7% (-0.4%, 1.8%)<br>0.4% (-0.4%, 1.2%)<br>0.3% (-0.3%, 0.9%)<br>0.1% (-1.1%, 1.3%) |
| Bowel obstruction; n (%) Gastroparesis; n (%) Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of SGLT-2; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformir, n (%) Past use of Insulins; n (%) | 167 (0.3%)<br>533 (0.8%)<br>219 (0.83)<br>200 [2.00, 3.00]<br>1.00, 6.00<br>36,599 (57.9%)<br>10,558 (16.7%)<br>20,522 (32.5%)<br>3,585 (5.7%)<br>4,172 (6.6%)<br>42,319 (67.0%)<br>14,679 (23.2%) | 36 (0.2%)<br>107 (0.7%)<br>2.32 (0.90)<br>2.00 [2.00, 3.00]<br>1.00, 6.00<br>7.195 (49.2%)<br>5.854 (40.0%)<br>3.386 (23.1%)<br>1.880 (12.8%)<br>975 (6.7%)<br>9.505 (64.9%)<br>7.460 (51.0%) | 0.0% (-0.1%, 0.1%)<br>0.1% (-0.0%, 0.3%)<br>-0.12 (-0.14, -0.11)<br>-(-,-)<br>-(-,-)<br>-(-,-)<br>8.8% (7.9%, 9.7%)<br>23.3% (-24.1%, -22.4%)<br>9.3% (8.6%, 10.1%)<br>-7.2% (-7.7%, -6.6%)<br>-0.1% (-0.5%, 0.4%)<br>2.0% (1.2%, 2.9%)<br>-27.7% (-28.6%, -26.9%) | 34 (0.3%)<br>89 (0.7%)<br>229 (0.89)<br>200 (2.00, 3.00)<br>1.00, 6.00<br>6.341 (51.4%)<br>4.156 (33.7%)<br>3.182 (25.8%)<br>1.408 (11.4%)<br>862 (7.0%)<br>8.183 (66.3%)<br>5.415 (43.9%) | 29 (0.2%)<br>89 (0.7%)<br>2.28 (0.89)<br>2.00 [2.00, 3.00]<br>1.00, 6.00<br>6.364 (51.6%)<br>4.126 (33.4%)<br>3.097 (25.1%)<br>1.361 (11.0%)<br>825 (6.7%)<br>8174 (66.2%)<br>5.377 (43.6%) | 0.0% (-0.1%, 0.2%)<br>0.0% (-0.2%, 0.2%)<br>0.01 (-0.01, 0.04)<br>-(-,-)<br>-(-,-)<br>-(-,-)<br>-0.2% (-1.4%, 1.1%)<br>0.2% (-0.9%, 1.4%)<br>0.7% (-0.4%, 1.8%)<br>0.4% (-0.4%, 1.2%)<br>0.3% (-0.3%, 0.9%)<br>0.1% (-1.1%, 1.3%)<br>0.3% (-0.9%, 1.6%) |
| Bowel obstruction; n (%) Gastroparesis; n (%) Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of SGLT-2t; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformin; n (%) Past use of Insulins; n (%) Past use of Sulfonylureas; n (%) | 167 (0.3%) 533 (0.8%) 219 (0.83) 200 [2.00, 3.00] 100, 6.00 36,599 (57.9%) 10,558 (16.7%) 20,522 (32.5%) 3,585 (5.7%) 4,172 (6.6%) 42,319 (67.0%) 14,679 (23.2%) 26,424 (41.8%) | 36 (0.2%)<br>107 (0.7%)<br>232 (0.90)<br>200 [2.00, 3.00]<br>1.00, 6.00<br>7.195 (49.2%)<br>5.854 (40.0%)<br>3.386 (23.1%)<br>1.880 (12.8%)<br>9.505 (64.9%)<br>7,460 (51.0%)<br>4,856 (33.2%) | 0.0% (-0.1%, 0.1%) 0.1% (-0.0%, 0.3%) -0.12 (-0.14, -0.11) -(·,-) -(·,-) 8.8% (7.9%, 9.7%) -2.3.3% (-24.1%, -22.4%) 9.3% (8.6%, 10.1%) -7.2% (-7.7%, -6.6%) -0.1% (-0.5%, 0.4%) 2.0% (1.2%, 2.9%) 2.77% (-28.6%, 26.9%) 8.6% (7.8%, 9.5%) | 34 (0.3%)<br>89 (0.7%)<br>229 (0.89)<br>200 (2.00, 3.00)<br>1.00, 6.00<br>6.341 (51.4%)<br>4,156 (33.7%)<br>3,182 (25.8%)<br>1,408 (11.4%)<br>862 (7.0%)<br>8,183 (66.3%)<br>5,415 (43.9%)<br>4,447 (36.0%) | 29 (0.2%)<br>89 (0.7%)<br>228 (0.89)<br>2.00 (2.00, 3.00)<br>1.00, 6.00<br>6.364 (51.6%)<br>4.126 (33.4%)<br>3.097 (25.1%)<br>1.361 (11.0%)<br>825 (6.7%)<br>8.174 (66.2%)<br>5.377 (43.6%)<br>4.337 (35.1%) | 0.0% (-0.1%, 0.2%)<br>0.0% (-0.2%, 0.2%)<br>0.01 (-0.01, 0.04)<br>-(;-)<br>-(;-)<br>-(;-)<br>-0.2% (-0.9%, 1.4%)<br>0.7% (-0.4%, 1.8%)<br>0.4% (-0.4%, 1.2%)<br>0.3% (-0.3%, 0.9%)<br>0.1% (-1.1%, 1.3%)<br>0.3% (-0.9%, 1.6%)<br>0.9% (-0.9%, 1.6%) |
| Bowel obstruction; n (%) Gastroparesis; n (%) Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of Solt-7: h n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Insulins; n (%) Past use of finsulins; n (%) Past use of Solt-7: h (%) | 167 (0.3%) 533 (0.8%) 219 (0.83) 2.00 [2.00, 3.00] 1.00, 6.00 36,599 (57.9%) 10,558 (16.7%) 20,522 (32.5%) 3,585 (5.7%) 41,72 (6.6%) 42,319 (67.0%) 14,679 (23.2%) 26,424 (41.8%) 5,619 (8.9%) 6,211 (9.8%) | 36 (0.2%)<br>107 (0.7%)<br>2.32 (0.90)<br>2.00 (2.00, 3.00)<br>1.00, 6.00<br>7.195 (49.2%)<br>5.854 (40.0%)<br>3.386 (23.1%)<br>1.880 (12.8%)<br>9.75 (6.7%)<br>9.505 (64.9%)<br>7.460 (51.0%)<br>4.856 (33.2%)<br>2.757 (18.8%)<br>1.568 (10.7%) | 0.0% (-0.1%, 0.1%) 0.1% (-0.0%, 0.3%) -0.12 (-0.14, -0.11) -(-, -) -(- | 34 (0.3%)<br>89 (0.7%)<br>229 (0.89)<br>200 (2.00, 3.00)<br>1.00, 6.00<br>6.341 (51.4%)<br>4.156 (33.7%)<br>3.182 (25.8%)<br>1,408 (11.4%)<br>862 (7.0%)<br>8.183 (66.3%)<br>5.415 (43.9%)<br>4.447 (36.0%)<br>2.061 (16.7%)<br>1,381 (11.2%) | 29 (0.2%)<br>89 (0.7%)<br>2.28 (0.89)<br>2.00 (2.00, 3.00)<br>1.00, 6.00<br>6.364 (51.6%)<br>4.126 (33.4%)<br>3.097 (25.1%)<br>1,361 (11.0%)<br>8.174 (66.2%)<br>5.377 (43.6%)<br>4.337 (35.1%)<br>2.018 (16.4%)<br>1,303 (10.6%) | 0.0% (-0.1%, 0.2%)<br>0.0% (-0.2%, 0.2%)<br>0.01 (-0.01, 0.04)<br>-(-, -)<br>-(-, - |
| Bowel obstruction; n (%) Gastroparesis; n (%) Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfornylureas; n (%) Concomitant use or initiation of Sulfornylureas; n (%) Concomitant use or initiation of Solf-Zi; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformir; n (%) Past use of Sulfornylureas; n (%) Past use of Sulfornylureas; n (%) Past use of Sulfornylureas; n (%) Past use of Sulfornylureas; n (%) Past use of Sulfornylureas; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) | 167 (0.3%) 533 (0.8%) 219 (0.83) 200 [2.00, 3.00] 1.00, 6.00 36,599 (57.9%) 10,558 (16.7%) 20,522 (32.5%) 3,585 (5.7%) 4,172 (6.6%) 42,319 (67.0%) 14,679 (23.2%) 26,424 (41.8%) 5,619 (8.9%) 6,211 (9.8%) 49,068 (77.7%) | 36 (0.2%)<br>107 (0.7%)<br>2.32 (0.90)<br>2.00 [2.00, 3.00]<br>1.00, 6.00<br>7.195 (49.2%)<br>5.854 (40.0%)<br>3.386 (23.1%)<br>1.880 (12.8%)<br>975 (6.7%)<br>9,505 (64.9%)<br>7.460 (51.0%)<br>4.856 (33.2%)<br>2.757 (18.8%)<br>1.568 (10.7%)<br>11,563 (79.0%) | 0.0% (-0.1%, 0.1%) 0.1% (-0.0%, 0.3%) -0.12 (-0.14, -0.11) -(·, -) -(·, -) -(·, -) 8.8% (7.9%, 9.7%) 23.3% (-24.1%, -22.4%) 9.3% (8.6%, 10.1%) -7.2% (-7.7%, -6.6%) -0.1% (-0.5%, 0.4%) 20% (1.2%, 2.9%) -27.7% (-28.6%, -26.9%) 8.6% (7.8%, 9.5%) -9.9% (-10.6%, -9.3%) -0.9% (-1.4%, -0.3%) -0.9% (-1.4%, -0.3%) | 34 (0.3%)<br>89 (0.7%)<br>2.29 (0.89)<br>2.00 [2.00, 3.00]<br>1.00, 6.00<br>6.341 (51.4%)<br>4.156 (33.7%)<br>3.182 (25.8%)<br>1.408 (11.4%)<br>862 (7.0%)<br>8.183 (66.3%)<br>5.415 (43.9%)<br>4.447 (36.0%)<br>2.061 (16.7%)<br>1.381 (11.2%)<br>9,764 (79.1%) | 29 (0.2%)<br>89 (0.7%)<br>2.28 (0.89)<br>2.00 [2.00, 3.00]<br>1.00, 6.00<br>6.364 (51.6%)<br>4.126 (33.4%)<br>3.097 (25.1%)<br>1.361 (11.0%)<br>825 (6.7%)<br>8.174 (66.2%)<br>5.377 (43.6%)<br>4,337 (35.1%)<br>2.018 (16.4%)<br>1.303 (10.6%)<br>9.678 (78.4%) | 0.0% (-0.1%, 0.2%)<br>0.0% (-0.2%, 0.2%)<br>0.01 (-0.01, 0.04)<br>-(·, -)<br>-(·, - |
| Bowel obstruction; n (%) Gastroparesis; n (%) Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of SGLT-2; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformin; n (%) Past use of Sulfonylureas; n (%) Past use of SicIT-2; n (%) Past use of SolT-7; n (%) Past use of Any other glucose-lowering drugs; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ARNI; n (%) | 167 (0.3%) 533 (0.8%) 219 (0.83) 200 [2.00, 3.00] 100, 6.00 36,599 (57.9%) 10,558 (16.7%) 20,522 (32.5%) 3,585 (5.7%) 4,172 (6.6%) 42,319 (67.0%) 14,679 (23.2%) 26,424 (41.8%) 5,619 (8.9%) 6,211 (9.8%) 49,068 (77.7%) 678 (1.1%) | 36 (0.2%)<br>107 (0.7%)<br>2.32 (0.90)<br>2.00 (2.00, 3.00)<br>1.00, 6.00<br>7.195 (49.2%)<br>5.854 (40.0%)<br>3.386 (23.1%)<br>1.880 (12.8%)<br>975 (6.7%)<br>9.505 (64.9%)<br>7.460 (51.0%)<br>4.856 (33.2%)<br>2.757 (18.8%)<br>1.568 (10.7%)<br>11.563 (79.0%)<br>213 (1.5%) | 0.0% (-0.1%, 0.1%) 0.1% (-0.0%, 0.3%) -0.12 (-0.14, -0.11) -(·,-) -(·,-) -(·,-) 8.8% (7.9%, 9.7%) 23.3% (-24.1%, -22.4%) 9.3% (8.6%, 10.1%) -7.2% (-7.7%, -6.6%) -0.1% (-0.5%, 0.4%) 2.0% (1.2%, 2.9%) 2.7% (-28.6%, -26.9%) 8.6% (7.8%, 9.5%) -9.9% (-10.6%, -9.3%) -0.9% (-1.4%, -0.3%) -1.4% (-2.1%, -0.6%) -0.4% (-0.6%, -0.2%) | 34 (0.3%)<br>89 (0.7%)<br>229 (0.89)<br>200 (2.00, 3.00)<br>1.00, 6.00<br>6.341 (51.4%)<br>4.156 (33.7%)<br>3.182 (25.8%)<br>1.408 (11.4%)<br>862 (7.0%)<br>8.183 (66.3%)<br>5.415 (43.9%)<br>4.447 (36.0%)<br>2061 (16.7%)<br>1,381 (112%)<br>9,764 (79.1%) | 29 (0.2%) 89 (0.7%) 228 (0.89) 2.00 (2.00, 3.00) 1.00, 6.00 6.364 (51.6%) 4,126 (33.4%) 3.097 (25.1%) 1.361 (11.0%) 825 (6.7%) 8,174 (66.2%) 5,377 (43.6%) 4,337 (35.1%) 2.018 (16.4%) 1,303 (10.6%) 9,678 (78.4%) 177 (1.4%) | 0.0% (-0.1%, 0.2%)<br>0.0% (-0.2%, 0.2%)<br>0.01 (-0.01, 0.04)<br>-(·, ·)<br>-(·, · |
| Bowel obstruction; n (%) Gastroparesis; n (%) Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of SULT-2i; n (%) Concomitant use or initiation of SULT-2i; n (%) Past use of Metformin; n (%) Past use of Insulins; n (%) Past use of Sulfonylureas; n (%) Past use of Sulfonylureas; n (%) Past use of Sulfonylureas; n (%) Past use of Any other glucose-lowering drugs; n (%) Past use of Sulfonylureas; n (%) | 167 (0.3%) 533 (0.8%) 219 (0.83) 200 [2.00, 3.00] 1.00, 6.00 36,599 (57.9%) 10,558 (16.7%) 20,522 (32.5%) 3,585 (5.7%) 4,172 (6.6%) 42,319 (67.0%) 14,679 (23.2%) 5,619 (8.9%) 6,211 (9.8%) 49,068 (77.7%) 678 (11%) 22,378 (35.4%) | 36 (0.2%) 107 (0.7%) 107 (0.7%) 2.32 (0.90) 2.00 (2.00, 3.00) 1.00, 6.00 7.195 (49.2%) 5.854 (40.0%) 3.386 (23.1%) 1.880 (12.8%) 9.505 (64.9%) 7.460 (51.0%) 4.856 (33.2%) 2.757 (18.8%) 1.568 (10.7%) 11,563 (79.0%) 213 (1.5%) 5.334 (36.4%) | 0.0% (-0.1%, 0.1%) 0.1% (-0.0%, 0.3%) -0.12 (-0.14, -0.11) -(.,-) -(.,-) -(.,-) -(.,-) -23.3% (-24.1%, -22.4%) 9.3% (8.6%, 10.1%) -7.2% (-7.7%, -6.6%) -0.1% (-0.5%, 0.4%) 2.0% (1.2%, 2.9%) 27.7% (-28.6%, -26.9%) 8.6% (-10.6%, -9.3%) -9.9% (-1.4%, -0.3%) -1.4% (-0.5%, 0.04%) -0.9% (-1.4%, -0.3%) -1.4% (-0.5%, 0.2%) | 34 (0.3%)<br>89 (0.7%)<br>2.29 (0.89)<br>2.00 (2.00, 3.00)<br>1.00, 6.00<br>6.341 (51.4%)<br>4.156 (33.7%)<br>3.182 (25.8%)<br>1.408 (11.4%)<br>862 (7.0%)<br>8.183 (66.3%)<br>5.415 (43.9%)<br>4.447 (36.0%)<br>2.061 (16.7%)<br>1.381 (11.2%)<br>9,764 (79.1%)<br>4.481 (36.3%) | 29 (0.2%) 89 (0.7%) 2.28 (0.89) 2.00 (2.00, 3.00) 1.00, 6.00 6.364 (61.6%) 4,126 (33.4%) 3,097 (25.1%) 1,361 (11.0%) 825 (6.7%) 8,174 (66.2%) 5,377 (43.6%) 4,373 (35.1%) 2,018 (16.4%) 1,303 (10.6%) 9,678 (78.4%) 1177 (1.4%) 4,473 (36.3%) | 0.0% (-0.1%, 0.2%)<br>0.0% (-0.2%, 0.2%)<br>0.01 (-0.01, 0.04)<br>-(·,·)<br>-( |
| Bowel obstruction; n (%) Gastroparesis; n (%) Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of SCLT-2; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Insulins; n (%) Past use of Sulfonylureas; n (%) Past use of Sulfonylureas; n (%) Past use of SaltT-2; n (%) Past use of SaltT-2; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ARN; n (%) Beta-blockers; n (%) Beta-blockers; n (%) | 167 (0.3%) 533 (0.8%) 219 (0.83) 2.00 [2.00, 3.00] 1.00, 6.00 36,599 (57.9%) 10,558 (16.7%) 20,522 (32.5%) 3,585 (5.7%) 4,172 (6.6%) 42,319 (67.0%) 14,679 (23.2%) 26,424 (41.8%) 5,619 (8.9%) 6,211 (9.8%) 49,068 (77.7%) 678 (1.1%) 22,378 (35.4%) 36,685 (58.1%) | 36 (0.2%) 107 (0.7%) 2.32 (0.90) 2.00 [2.00, 3.00] 1.00, 6.00 7.195 (49.2%) 5.854 (40.0%) 3.386 (23.1%) 1.880 (12.8%) 9.505 (64.9%) 7.460 (51.0%) 4.856 (33.2%) 2.757 (18.8%) 1.568 (10.7%) 11.563 (79.0%) 213 (1.5%) 5.334 (36.4%) 8.676 (59.3%) | 0.0% (-0.1%, 0.1%) 0.1% (-0.0%, 0.3%) -0.12 (-0.14, -0.11) -(-, -) -(- | 34 (0.3%)<br>89 (0.7%)<br>2.29 (0.89)<br>2.00 [2.00, 3.00]<br>1.00, 6.00<br>6.341 (51.4%)<br>4,156 (33.7%)<br>3,182 (25.8%)<br>1,408 (11.4%)<br>962 (7.0%)<br>8,183 (66.3%)<br>5,415 (43.9%)<br>4,447 (36.0%)<br>2,061 (16.7%)<br>1,381 (11.2%)<br>9,764 (79.1%)<br>154 (1.2%)<br>4,481 (36.3%)<br>7,143 (57.9%) | 29 (0.2%) 89 (0.7%) 2.28 (0.89) 2.00 (2.00, 3.00) 1.00, 6.00 6.364 (51.6%) 4.126 (33.4%) 3.097 (25.1%) 1.361 (11.0%) 825 (6.7%) 8.174 (66.2%) 5.377 (43.6%) 4.337 (35.1%) 2.018 (16.4%) 1,303 (10.6%) 9.678 (78.4%) 177 (1.4%) 4.473 (36.3%) 7,158 (58.0%) | 0.0% (-0.1%, 0.2%) 0.0% (-0.2%, 0.2%) 0.01 (-0.01, 0.04) -(-, -) -(-, |
| Bowel obstruction; n (%) Gastroparesis; n (%) Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfornylureas; n (%) Concomitant use or initiation of Sulfornylureas; n (%) Concomitant use or initiation of Sulfornylureas; n (%) Concomitant use or initiation of Solt-Zi; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformin; n (%) Past use of Sulfornylureas; n (%) Past use of Sulfornylureas; n (%) Past use of Sulfornylureas; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ARN; n (%) Beta-blockers; n (%) Calcium channel blockers; n (%) | 167 (0.3%) 533 (0.8%) 219 (0.83) 200 [2.00, 3.00] 1.00, 6.00 36,599 (57.9%) 10,558 (16.7%) 20,522 (32.5%) 3,585 (5.7%) 4,172 (6.6%) 42,319 (67.0%) 14,679 (23.2%) 26,424 (41.8%) 5,619 (8.9%) 6,211 (9.8%) 49,068 (77.7%) 678 (1.1%) 22,378 (35.4%) 36,685 (58.1%) 25,814 (40.9%) | 36 (0.2%) 107 (0.7%) 2.32 (0.90) 2.00 [2.00, 3.00] 1.00, 6.00 7,195 (49.2%) 5.854 (40.0%) 3,386 (23.1%) 1,880 (12.8%) 975 (6.7%) 9,505 (64.9%) 7,460 (51.0%) 4,856 (33.2%) 2,757 (18.8%) 1,568 (10.7%) 11,563 (79.0%) 213 (1.5%) 5,334 (36.4%) 8,676 (59.3%) 5,554 (38.0%) | 0.0% (-0.1%, 0.1%) 0.1% (-0.0%, 0.3%) -0.12 (-0.14, -0.11) -(-,-) -(-,-) -(-,-) 8.8% (7.9%, 9.7%) 23.3% (224.1%, -22.4%) 9.3% (8.6%, 10.1%) 7.2% (-7.7%, -6.6%) -0.1% (-0.5%, 0.4%) 20% (1.2%, 2.9%) -27.7% (-28.6%, -26.9%) 8.6% (7.8%, 9.5%) -9.9% (-10.6%, -9.3%) -9.9% (-10.6%, -0.3%) -1.4% (-2.1%, -0.6%) -0.4% (-0.6%, -0.2%) -1.0% (-1.9%, -0.2%) -1.2% (-2.1%, -0.3%) 2.9% (2.0%, 3.8%) | 34 (0.3%)<br>89 (0.7%)<br>2.29 (0.89)<br>2.00 (2.00, 3.00)<br>1.00, 6.00<br>6.341 (51.4%)<br>4.156 (33.7%)<br>3.182 (25.8%)<br>1.408 (11.4%)<br>862 (7.0%)<br>8.183 (66.3%)<br>5.415 (43.9%)<br>4.447 (36.0%)<br>2.061 (16.7%)<br>1.381 (11.2%)<br>9.764 (79.1%)<br>154 (1.2%)<br>4.481 (36.3%)<br>7.143 (57.9%)<br>4.722 (38.3%) | 29 (0.2%) 89 (0.7%) 228 (0.89) 2.00 [2.00, 3.00] 1.00, 6.00 6.364 (51.6%) 4,126 (33.4%) 3.097 (25.1%) 1.361 (11.0%) 825 (6.7%) 8,174 (66.2%) 5,377 (43.6%) 4,337 (35.1%) 2,018 (16.4%) 1,303 (10.6%) 9,678 (78.4%) 177 (1.4%) 4,473 (36.3%) 7,1518 (58.0%) 4,705 (38.1%) | 0.0% (-0.1%, 0.2%) 0.0% (-0.2%, 0.2%) 0.01 (-0.01, 0.04) -(·,-) -(·,-) -(·,-) -(·,-) -(·,-) -(·,-) 0.2% (-1.4%, 1.1%) 0.2% (-0.9%, 1.4%) 0.7% (-0.4%, 1.8%) 0.4% (-0.4%, 1.2%) 0.3% (-0.3%, 0.9%) 0.1% (-1.1%, 1.3%) 0.3% (-0.9%, 1.6%) 0.9% (-0.3%, 2.1%) 0.3% (-0.9%, 1.6%) 0.3% (-0.9%, 1.6%) 0.3% (-0.9%, 1.6%) 0.3% (-0.9%, 1.6%) 0.3% (-0.9%, 1.3%) 0.3% (-0.9%, 1.3%) 0.3% (-0.9%, 1.3%) 0.1% (-1.1%, 1.3%) 0.1% (-1.1%, 1.3%) 0.1% (-1.1%, 1.4%) |
| Bowel obstruction; n (%) Gastroparesis; n (%) Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of SGLT-2; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformin; n (%) Past use of Sulfonylureas; n (%) Past use of Sulfonylureas; n (%) Past use of SGLT-2; n (%) Past use of Any other glucose-lowering drugs; n (%) ARNI; n (%) Thiazides; n (%) Beta-blockers; n (%) Beta-blockers; n (%) Digoxin / Digitoxin; n (%) | 167 (0.3%) 533 (0.8%) 219 (0.83) 2.00 [2.00, 3.00] 1.00, 6.00 36,599 (57.9%) 10,558 (16.7%) 20,522 (32.5%) 4,172 (6.6%) 42,319 (67.0%) 14,679 (23.2%) 56,619 (8.9%) 6,211 (9.8%) 49,068 (77.7%) 678 (1.1%) 22,378 (35.4%) 36,685 (58.1%) 25,814 (40.9%) 1,667 (2.6%) | 36 (0.2%) 107 (0.7%) 107 (0.7%) 2.32 (0.90) 2.00 (2.00, 3.00) 1.00, 6.00 7.195 (49.2%) 5.854 (40.0%) 3.386 (23.1%) 1.880 (12.8%) 975 (6.7%) 9.505 (64.9%) 7.460 (51.0%) 4.856 (33.2%) 2.757 (18.8%) 1.568 (10.7%) 11.563 (79.0%) 213 (1.5%) 5.334 (36.4%) 8.676 (59.3%) 5.554 (38.0%) 309 (2.1%) | 0.0% (-0.1%, 0.1%) 0.1% (-0.0%, 0.3%) 0.12 (-0.14, -0.11) -(-,-) | 34 (0.3%)<br>89 (0.7%)<br>229 (0.89)<br>200 (2.00, 3.00)<br>1.00, 6.00<br>6.341 (51.4%)<br>4.156 (33.7%)<br>3.182 (25.8%)<br>1.408 (11.4%)<br>862 (7.0%)<br>8.183 (66.3%)<br>5.415 (43.9%)<br>4.447 (36.0%)<br>2.061 (16.7%)<br>1.381 (11.2%)<br>9.764 (79.1%)<br>154 (12.3%)<br>4.481 (36.3%)<br>7.143 (57.9%)<br>4.722 (38.3%)<br>244 (2.0%) | 29 (0.2%) 89 (0.7%) 2.28 (0.89) 2.00 (2.00, 3.00) 1.00, 6.00 6.364 (61.6%) 4,126 (33.4%) 3,097 (25.1%) 1,361 (11.0%) 825 (6.7%) 8,174 (66.2%) 5,377 (43.6%) 4,337 (35.1%) 2,018 (16.4%) 1,303 (10.6%) 9,678 (78.4%) 1,77 (1.4%) 4,473 (36.3%) 7,158 (58.0%) 4,705 (38.1%) 262 (2.1%) | 0.0% (-0.1%, 0.2%)<br>0.0% (-0.2%, 0.2%)<br>0.01 (-0.01, 0.04)<br>-(-, -)<br>-(-, -)<br>-0.2% (-0.9%, 1.4%)<br>0.2% (-0.9%, 1.4%)<br>0.7% (-0.4%, 1.8%)<br>0.3% (-0.3%, 0.9%)<br>0.3% (-0.3%, 0.9%)<br>0.3% (-0.3%, 0.9%)<br>0.3% (-0.6%, 1.3%)<br>0.5% (-0.3%, 1.7%)<br>0.5% (-0.3%, 1.7%)<br>0.5% (-0.3%, 1.7%)<br>0.1% (-1.1%, 1.3%)<br>0.1% (-0.5%, 0.1%)<br>0.1% (-1.1%, 1.3%)<br>0.1% (-1.1%, 1.3%) |
| Bowel obstruction; n (%) Gastroparesis; n (%) Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of SGLT-2i; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformin; n (%) Past use of Insulins; n (%) Past use of Sulfonylureas; n (%) Past use of Sulfonylureas; n (%) Past use of Any other glucose-lowering drugs; n (%) Past use of Any other glucose-lowering drugs; n (%) Past use of Insulins; n (%) Past use of Self-2i; n (%) Past use of Insulins; n (%) Past use of Self-7i; n (%) Past use of Insulins; n | 167 (0.3%) 533 (0.8%) 219 (0.83) 2.00 [2.00, 3.00] 1.00, 6.00 36,599 (57.9%) 10,558 (16.7%) 20,522 (32.5%) 3.585 (5.7%) 41,72 (6.6%) 42,319 (67.0%) 14,679 (23.2%) 26,424 (41.8%) 5,619 (8.9%) 6,211 (9.8%) 49,068 (77.7%) 678 (11%) 22,378 (35.4%) 36,685 (58.1%) 25,814 (40.9%) 1,667 (2.6%) 20,432 (32.3%) | 36 (0.2%) 107 (0.7%) 107 (0.7%) 2.32 (0.90) 2.00 [2.00, 3.00] 1.00, 6.00 7.195 (49.2%) 5.854 (40.0%) 3.386 (23.1%) 1.880 (12.8%) 9.505 (64.9%) 7.460 (51.0%) 4.856 (33.2%) 2.757 (18.8%) 1.568 (10.7%) 11,563 (79.0%) 213 (1.5%) 5.334 (36.4%) 8.676 (59.3%) 5.554 (38.0%) 3.99 (21%) 5.125 (35.0%) | 0.0% (-0.1%, 0.1%) 0.1% (-0.0%, 0.3%) -0.12 (-0.14, -0.11) -(-, -) -( | 34 (0.3%) 89 (0.7%) 229 (0.89) 200 (2.00, 3.00) 1.00, 6.00 6.341 (51.4%) 4.156 (33.7%) 3.182 (25.8%) 1,408 (11.4%) 862 (7.0%) 8.183 (66.3%) 5.415 (43.9%) 4.447 (36.0%) 2.061 (16.7%) 1.381 (112%) 9,764 (79.1%) 154 (1.2%) 4,481 (36.3%) 7,143 (57.9%) 4,722 (38.3%) 4,722 (38.3%) 4,724 (2.0%) 4,140 (33.6%) | 29 (0.2%) 89 (0.7%) 228 (0.89) 2.00 (2.00, 3.00) 1.00, 6.00 6.364 (51.6%) 4,126 (33.4%) 3,097 (25.1%) 1,361 (11.0%) 825 (6.7%) 8,174 (66.2%) 5,377 (43.6%) 4,337 (35.1%) 2,018 (16.4%) 1,303 (10.6%) 9,678 (78.4%) 1,77 (1.4%) 4,473 (36.3%) 4,705 (38.1%) 262 (2.1%) 4,101 (33.2%) | 0.0% (-0.1%, 0.2%) 0.0% (-0.1%, 0.2%) 0.01 (-0.01, 0.04) -(·,·) - |
| Bowel obstruction; n (%) Gastroparesis; n (%) Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of SCLT-2; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Insulins; n (%) Past use of Insulins; n (%) Past use of Sulfonylureas; n (%) Past use of Sulfonylureas; n (%) Past use of Sulfonylureas; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ARN; n (%) Beta-blockers; n (%) Calcium channel blockers; n (%) Digoxin / Digitoxin; n (%) Loop diuretics; n (%) Other diuretics; n (%) Other diuretics; n (%) | 167 (0.3%) 533 (0.8%) 219 (0.83) 2.00 [2.00, 3.00] 1.00, 6.00 36,599 (57.9%) 10,558 (16.7%) 20,522 (32.5%) 3,585 (5.7%) 4,172 (6.6%) 42,319 (67.0%) 14,679 (23.2%) 26,424 (41.8%) 5,619 (8.9%) 6,211 (9.8%) 49,068 (77.7%) 678 (1.1%) 22,378 (35.4%) 36,685 (58.1%) 25,814 (40.9%) 1,667 (2.6%) 1,667 (2.6%) 6,557 (10.4%) | 36 (0.2%) 107 (0.7%) 2.32 (0.90) 2.00 [2.00, 3.00] 1.00, 6.00 7.195 (49.2%) 5.854 (40.0%) 3.386 (23.1%) 1.880 (12.8%) 9.505 (64.9%) 7.460 (51.0%) 4.856 (33.2%) 2.757 (18.8%) 1.568 (10.7%) 11,563 (79.0%) 213 (1.5%) 5.334 (36.4%) 8.676 (59.3%) 5.554 (38.0%) 309 (21%) 5.125 (35.0%) 1.888 (12.6%) | 0.0% (-0.1%, 0.1%) 0.1% (-0.0%, 0.3%) -0.12 (-0.14, -0.11) -(-, -) -(- | 34 (0.3%) 89 (0.7%) 229 (0.89) 2.00 [2.00, 3.00] 1.00, 6.00 6.341 (51.4%) 4,156 (33.7%) 3,182 (25.8%) 1,408 (11.4%) 962 (7.0%) 8,183 (66.3%) 5,415 (43.9%) 4,447 (36.0%) 2,061 (16.7%) 1,381 (11.2%) 9,764 (79.1%) 154 (1.2%) 4,481 (36.3%) 7,143 (57.9%) 4,722 (38.3%) 244 (2.0%) 4,140 (33.6%) 1,458 (11.8%) | 29 (0.2%) 89 (0.7%) 228 (0.89) 2.00 (2.00, 3.00) 1.00, 6.00 6.364 (51.6%) 4,126 (33.4%) 3.097 (25.1%) 1,361 (11.0%) 8174 (66.2%) 5.377 (43.6%) 4,337 (35.1%) 2.018 (16.4%) 1,303 (10.6%) 9,678 (78.4%) 177 (1.4%) 4,473 (36.3%) 7,158 (58.0%) 4,705 (38.1%) 262 (2.1%) 4,101 (33.2%) 1,437 (11.6%) | 0.0% (-0.1%, 0.2%) 0.0% (-0.1%, 0.2%) 0.01 (-0.01, 0.04) -(-, -) -(-, |
| Bowel obstruction; n (%) Gastroparesis; n (%) Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfornylureas; n (%) Concomitant use or initiation of Sulfornylureas; n (%) Concomitant use or initiation of Sulfornylureas; n (%) Concomitant use or initiation of SQLT-2k n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformin; n (%) Past use of Sulfornylureas; n (%) Past use of Sulfornylureas; n (%) Past use of Sulfornylureas; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ARN; n (%) Thiazides; n (%) Calcium channel blockers; n (%) Calcium channel blockers; n (%) Upgoxin / Digitoxin; n (%) Loop diuretics; n (%) Intravenous diuretics; n (%) | 167 (0.3%) 533 (0.8%) 219 (0.83) 200 [2.00, 3.00] 1.00, 6.00 36,599 (57.9%) 10,558 (16.7%) 20,522 (32.5%) 3,585 (5.7%) 4,172 (6.6%) 42,319 (67.0%) 14,679 (23.2%) 26,424 (41.8%) 5,619 (8.9%) 6,211 (9.8%) 49,068 (77.7%) 678 (1.1%) 22,378 (35.4%) 36,685 (58.1%) 25,814 (40.9%) 1,667 (2.6%) 20,432 (32.3%) 6,557 (10.4%) 1,769 (2.8%) | 36 (0.2%) 107 (0.7%) 2.32 (0.90) 2.00 [2.00, 3.00] 1.00, 6.00 7.195 (49.2%) 5.854 (40.0%) 3.386 (23.1%) 1.880 (12.8%) 975 (6.7%) 9,505 (64.9%) 7.460 (51.0%) 4.856 (33.2%) 2.757 (18.8%) 11.563 (79.0%) 213 (1.5%) 5.334 (36.4%) 8.676 (59.3%) 5.554 (38.0%) 309 (21%) 5.125 (35.0%) 1.838 (12.6%) 384 (2.6%) | 0.0% (-0.1%, 0.1%) 0.1% (-0.0%, 0.3%) -0.12 (-0.14, -0.11) -(-, -) -( | 34 (0.3%) 89 (0.7%) 229 (0.89) 2.00 [2.00, 3.00] 1.00, 6.00 6.341 (51.4%) 4.156 (33.7%) 3.182 (25.8%) 1.408 (11.4%) 862 (7.0%) 8.183 (66.3%) 5.415 (43.9%) 4.447 (36.0%) 2.061 (16.7%) 1.381 (11.2%) 9.764 (79.1%) 154 (1.2%) 4.481 (36.3%) 7.143 (57.9%) 4.722 (38.3%) 244 (20%) 4.140 (33.6%) 1.458 (11.8%) 312 (25.%) | 29 (0.2%) 89 (0.7%) 228 (0.89) 2.00 [2.00, 3.00] 1.00, 6.00 6.364 (51.6%) 4,126 (33.4%) 3,097 (25.1%) 1.361 (11.0%) 825 (6.7%) 8,174 (66.2%) 5,377 (43.6%) 4,337 (35.1%) 2,018 (16.4%) 1,303 (10.6%) 9,678 (78.4%) 177 (1.4%) 4,473 (36.3%) 7,756 (38.1%) 262 (21%) 4,101 (33.2%) 1,437 (11.6%) 311 (2.5%) | 0.0% (-0.1%, 0.2%) 0.0% (-0.1%, 0.2%) 0.0% (-0.2%, 0.2%) 0.01 (-0.01, 0.04) -(-, -) -( |
| Bowel obstruction; n (%) Gastroparesis; n (%) Number of antidiabetic drugs on CEDmean (sd)median (IQR)min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of SGLT-2; n (%) Concomitant use or initiation of SGLT-2; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformin; n (%) Past use of Insulins; n (%) Past use of Sulfonylureas; n (%) Past use of Sulfonylureas; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ACE-is/ARB's; n (%) STIPLIAND (SM) ST | 167 (0.3%) 533 (0.8%) 219 (0.83) 200 [2.00, 3.00] 1.00, 6.00 36,599 (57.9%) 10,558 (16.7%) 20,522 (32.5%) 3,585 (5.7%) 4,172 (6.6%) 42,319 (67.0%) 14,679 (23.2%) 5,619 (8.9%) 6,211 (9.8%) 49,068 (77.7%) 678 (1.1%) 22,378 (35.4%) 36,685 (58.1%) 22,378 (35.4%) 36,685 (58.1%) 20,432 (32.3%) 6,557 (10.4%) 1,769 (2.6%) | 36 (0.2%) 107 (0.7%) 107 (0.7%) 2.32 (0.90) 2.00 (2.00, 3.00) 1.00, 6.00 7.195 (49.2%) 5.854 (40.0%) 3.386 (23.1%) 1.880 (12.8%) 975 (6.7%) 9.505 (64.9%) 7.460 (51.0%) 4.856 (33.2%) 2.757 (18.8%) 1.568 (10.7%) 11,563 (79.0%) 213 (1.5%) 5.334 (36.4%) 8.676 (59.3%) 5.554 (38.0%) 309 (2.1%) 5.125 (35.0%) 1.838 (12.6%) 1.838 (12.6%) 1.838 (12.6%) 1.995 (13.6%) | 0.0% (-0.1%, 0.1%) 0.1% (-0.0%, 0.3%) 0.12 (-0.14, -0.11) -(-, -) -(-, | 34 (0.3%) 89 (0.7%) 229 (0.89) 2.00 (2.00, 3.00) 1.00, 6.00 6.341 (51.4%) 4.156 (33.7%) 3.182 (25.8%) 1.408 (11.4%) 862 (7.0%) 8.183 (66.3%) 5.415 (43.9%) 4.447 (36.0%) 2.061 (16.7%) 1.381 (11.2%) 9,764 (79.1%) 154 (1.2%) 4.481 (36.3%) 7.143 (57.9%) 4.481 (36.3%) 7.143 (57.9%) 4.472 (38.3%) 244 (2.0%) 4.140 (33.6%) 1.458 (11.8%) 1.612 (13.1%) | 29 (0.2%) 89 (0.7%) 228 (0.89) 2.00 (2.00, 3.00) 1.00, 6.00 6.364 (51.6%) 4,126 (33.4%) 3,0.97 (25.1%) 1,361 (11.0%) 825 (6.7%) 8,174 (66.2%) 5,377 (43.6%) 4,337 (35.1%) 2,018 (16.4%) 1,303 (10.6%) 9,678 (78.4%) 177 (1.4%) 4,473 (36.3%) 4,473 (36.3%) 7,158 (58.0%) 4,705 (38.1%) 262 (2.1%) 4,101 (33.2%) 1,437 (11.6%) 311 (2.5%) 1,605 (13.0%) | 0.0% (-0.1%, 0.2%) 0.0% (-0.1%, 0.2%) 0.01 (-0.01, 0.04) -(·, ·) -(·, |
| Bowel obstruction; n (%) Gastroparesis; n (%) Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfornylureas; n (%) Concomitant use or initiation of Sulfornylureas; n (%) Concomitant use or initiation of Sulfornylureas; n (%) Concomitant use or initiation of SQLT-2k n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformin; n (%) Past use of Sulfornylureas; n (%) Past use of Sulfornylureas; n (%) Past use of Sulfornylureas; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ARN; n (%) Thiazides; n (%) Calcium channel blockers; n (%) Calcium channel blockers; n (%) Upgoxin / Digitoxin; n (%) Loop diuretics; n (%) Intravenous diuretics; n (%) | 167 (0.3%) 533 (0.8%) 219 (0.83) 2.00 [2.00, 3.00] 1.00, 6.00 36,599 (57.9%) 10,558 (16.7%) 20,522 (32.5%) 3,585 (5.7%) 41,72 (6.6%) 42,319 (67.0%) 14,679 (23.2%) 26,424 (41.8%) 5,619 (8.9%) 6,211 (9.8%) 49,068 (77.7%) 678 (11%) 22,378 (35.4%) 36,685 (58.1%) 25,814 (40.9%) 1,667 (2.6%) 20,432 (32.3%) 6,557 (10.4%) 1,769 (2.8%) 7,852 (12.4%) 2921 (4.6%) | 36 (0.2%) 107 (0.7%) 107 (0.7%) 2.32 (0.90) 2.00 [2.00, 3.00] 1.00, 6.00 7.195 (49.2%) 5.854 (40.0%) 3.386 (23.1%) 1.880 (12.8%) 9.505 (64.9%) 7.460 (51.0%) 4.856 (33.2%) 2.757 (18.8%) 1,568 (10.7%) 11,563 (79.0%) 1,563 (79.0%) 1,564 (38.0%) 3,34 (36.4%) 8,676 (59.3%) 5,554 (38.0%) 3,92 (21%) 5,125 (38.0%) 3,125 (38.0%) 3,126 (38.0%) | 0.0% (-0.1%, 0.1%) 0.1% (-0.0%, 0.3%) 0.12 (-0.14, -0.11) -(.,-) | 34 (0.3%) 89 (0.7%) 229 (0.89) 200 (2.00, 3.00) 1.00, 6.00 6.341 (51.4%) 4.156 (33.7%) 3.182 (25.8%) 1,408 (11.4%) 862 (7.0%) 8.183 (66.3%) 5.415 (43.9%) 4.447 (36.0%) 2.061 (16.7%) 1,381 (11.2%) 9,764 (79.1%) 154 (1.2%) 4,481 (36.3%) 7,143 (57.9%) 4,722 (38.3%) 244 (2.0%) 4,140 (33.6%) 1,458 (11.8%) 312 (2.5%) 1,612 (13.1%) 540 (4.4%) | 29 (0.2%) 89 (0.7%) 228 (0.89) 2.00 (2.00, 3.00) 1.00, 6.00 6.364 (51.6%) 4.126 (33.4%) 3.097 (25.1%) 1.361 (11.0%) 825 (6.7%) 8.174 (66.2%) 5.377 (43.6%) 4.337 (35.1%) 2.018 (16.4%) 1.303 (10.6%) 9,678 (78.4%) 1.77 (1.4%) 4.473 (36.3%) 7.158 (58.0%) 4,705 (38.1%) 262 (2.1%) 4,101 (33.2%) 1.437 (11.6%) 311 (2.5%) 1.605 (13.0%) 525 (4.3%) | 0.0% (-0.1%, 0.2%) 0.0% (-0.1%, 0.2%) 0.0% (-0.2%, 0.2%) 0.01 (-0.01, 0.04) -(·,·) -(· |
| Bowel obstruction; n (%) Gastroparesis; n (%) Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of SGLT-2; n (%) Concomitant use or initiation of SGLT-2; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformin; n (%) Past use of Insulins; n (%) Past use of Sulfonylureas; n (%) Past use of Sulfonylureas; n (%) Past use of Any other glucose-lowering drugs; n (%) Past use of Any other glucose-lowering drugs; n (%) Past use of Nover of the glucose-lowering drugs; n (%) Past use of Topic (%) Past use of Nover (%) Past use of Nover (%) Past use of Nover (%) Past use of Sulfonylureas; n (%) Past use of Topic (%) Past use of Topic (%) Past use of Topic (%) Past (%) | 167 (0.3%) 533 (0.8%) 219 (0.83) 200 [2.00, 3.00] 1.00, 6.00 36,599 (57.9%) 10,558 (16.7%) 20,522 (32.5%) 3,585 (5.7%) 4,172 (6.6%) 42,319 (67.0%) 14,679 (23.2%) 5,619 (8.9%) 6,211 (9.8%) 49,068 (77.7%) 678 (1.1%) 22,378 (35.4%) 36,685 (58.1%) 22,378 (35.4%) 36,685 (58.1%) 20,432 (32.3%) 6,557 (10.4%) 1,769 (2.6%) | 36 (0.2%) 107 (0.7%) 107 (0.7%) 2.32 (0.90) 2.00 (2.00, 3.00) 1.00, 6.00 7.195 (49.2%) 5.854 (40.0%) 3.386 (23.1%) 1.880 (12.8%) 975 (6.7%) 9.505 (64.9%) 7.460 (51.0%) 4.856 (33.2%) 2.757 (18.8%) 1.568 (10.7%) 11,563 (79.0%) 213 (1.5%) 5.334 (36.4%) 8.676 (59.3%) 5.554 (38.0%) 309 (2.1%) 5.125 (35.0%) 1.838 (12.6%) 1.838 (12.6%) 1.838 (12.6%) 1.995 (13.6%) | 0.0% (-0.1%, 0.1%) 0.1% (-0.0%, 0.3%) 0.12 (-0.14, -0.11) -(-, -) -(-, | 34 (0.3%) 89 (0.7%) 229 (0.89) 2.00 (2.00, 3.00) 1.00, 6.00 6.341 (51.4%) 4.156 (33.7%) 3.182 (25.8%) 1.408 (11.4%) 862 (7.0%) 8.183 (66.3%) 5.415 (43.9%) 4.447 (36.0%) 2.061 (16.7%) 1.381 (11.2%) 9,764 (79.1%) 154 (1.2%) 4.481 (36.3%) 7.143 (57.9%) 4.481 (36.3%) 7.143 (57.9%) 4.472 (38.3%) 244 (2.0%) 4.140 (33.6%) 1.458 (11.8%) 1.612 (13.1%) | 29 (0.2%) 89 (0.7%) 228 (0.89) 2.00 (2.00, 3.00) 1.00, 6.00 6.364 (51.6%) 4,126 (33.4%) 3,0.97 (25.1%) 1,361 (11.0%) 825 (6.7%) 8,174 (66.2%) 5,377 (43.6%) 4,337 (35.1%) 2,018 (16.4%) 1,303 (10.6%) 9,678 (78.4%) 177 (1.4%) 4,473 (36.3%) 4,473 (36.3%) 7,158 (58.0%) 4,705 (38.1%) 262 (2.1%) 4,101 (33.2%) 1,437 (11.6%) 311 (2.5%) 1,605 (13.0%) | 0.0% (-0.1%, 0.2%) 0.0% (-0.1%, 0.2%) 0.01 (-0.01, 0.04) -(·, ·) -(·, |
| Bowel obstruction; n (%) Gastroparesis; n (%) Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of SGLT-2!; n (%) Concomitant use or initiation of SGLT-2!; n (%) Concomitant use or initiation of SGLT-2!; n (%) Past use of Metformin; n (%) Past use of Insulins; n (%) Past use of Insulins; n (%) Past use of SGLT-2; n (%) Past use of SGLT-2; n (%) Past use of SGLT-3; n (%) Past use of SGLT-3; n (%) Past use of SGLT-3; n (%) Past use of Any other glucose-lowering drugs; n (%) Past use of Any other glucose-lowering drugs; n (%) Past use of Any other glucose-lowering drugs; n (%) Calcium channel blockers; n (%) Digoxin / Digitoxin; n (%) Loop diuretics; n (%) Intravenous diuretics; n (%) Anti-arrhythmics; n (%) | 167 (0.3%) 533 (0.8%) 219 (0.83) 2.00 [2.00, 3.00] 1.00, 6.00 36,599 (57.9%) 10,558 (16.7%) 20,522 (32.5%) 3,585 (5.7%) 41,72 (6.6%) 42,319 (67.0%) 14,679 (23.2%) 26,424 (41.8%) 5,619 (8.9%) 6,211 (9.8%) 49,068 (77.7%) 678 (11%) 22,378 (35.4%) 36,685 (58.1%) 25,814 (40.9%) 1,667 (2.6%) 20,432 (32.3%) 6,557 (10.4%) 1,769 (2.8%) 7,852 (12.4%) 2921 (4.6%) | 36 (0.2%) 107 (0.7%) 107 (0.7%) 2.32 (0.90) 2.00 [2.00, 3.00] 1.00, 6.00 7.195 (49.2%) 5.854 (40.0%) 3.386 (23.1%) 1.880 (12.8%) 9.505 (64.9%) 7.460 (51.0%) 4.856 (33.2%) 2.757 (18.8%) 1,568 (10.7%) 11,563 (79.0%) 1,563 (79.0%) 1,564 (38.0%) 3,34 (36.4%) 8,676 (59.3%) 5,554 (38.0%) 3,92 (21%) 5,125 (38.0%) 3,125 (38.0%) 3,126 (38.0%) | 0.0% (-0.1%, 0.1%) 0.1% (-0.0%, 0.3%) 0.12 (-0.14, -0.11) -(.,-) | 34 (0.3%) 89 (0.7%) 229 (0.89) 200 (2.00, 3.00) 1.00, 6.00 6.341 (51.4%) 4.156 (33.7%) 3.182 (25.8%) 1,408 (11.4%) 862 (7.0%) 8.183 (66.3%) 5.415 (43.9%) 4.447 (36.0%) 2.061 (16.7%) 1,381 (11.2%) 9,764 (79.1%) 154 (1.2%) 4,481 (36.3%) 7,143 (57.9%) 4,722 (38.3%) 244 (2.0%) 4,140 (33.6%) 1,458 (11.8%) 312 (2.5%) 1,612 (13.1%) 540 (4.4%) | 29 (0.2%) 89 (0.7%) 228 (0.89) 2.00 (2.00, 3.00) 1.00, 6.00 6.364 (51.6%) 4.126 (33.4%) 3.097 (25.1%) 1.361 (11.0%) 825 (6.7%) 8.174 (66.2%) 5.377 (43.6%) 4.337 (35.1%) 2.018 (16.4%) 1.303 (10.6%) 9,678 (78.4%) 1.77 (1.4%) 4.473 (36.3%) 7.158 (58.0%) 4,705 (38.1%) 262 (2.1%) 4,101 (33.2%) 1.437 (11.6%) 311 (2.5%) 1.605 (13.0%) 525 (4.3%) | 0.0% (-0.1%, 0.2%) 0.0% (-0.1%, 0.2%) 0.0% (-0.2%, 0.2%) 0.01 (-0.01, 0.04) -(·,·) -(· |
| Bowel obstruction; n (%) Gastroparesis; n (%) Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of SASLT-2i; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformin; n (%) Past use of Insulins; n (%) Past use of Sulfonylureas; n (%) Past use of Sulfonylureas; n (%) Past use of Sulfonylureas; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ARNI; n (%) Thiazides; n (%) Calcium channel blockers; n (%) Calcium channel blockers; n (%) Calcium channel blockers; n (%) Upop diuretics; n (%) Intravenous diuretics; n (%) Intravenous diuretics; n (%) Nitrates; n (%) PCSK9 inhibitors and other lipid-lowering drugs; n (%) | 167 (0.3%) 533 (0.8%) 219 (0.83) 200 [2.00, 3.00] 1.00, 6.00 36,599 (57.9%) 10,558 (16.7%) 20,522 (32.5%) 3,585 (5.7%) 4,172 (6.6%) 42,319 (67.0%) 14,679 (23.2%) 26,424 (41.8%) 5,619 (8.9%) 6,211 (9.8%) 49,068 (77.7%) 678 (1.1%) 22,378 (35.4%) 36,685 (58.1%) 25,814 (40.9%) 1,667 (2.6%) 20,432 (32.3%) 6,557 (10.4%) 1,769 (2.8%) 7,852 (12.4%) 2,921 (4.6%) 5,1100 (80.9%) 8,635 (13.7%) | 36 (0.2%) 107 (0.7%) 2.32 (0.90) 2.00 [2.00, 3.00] 1.00, 6.00 7.195 (49.2%) 5.854 (40.0%) 3.386 (23.1%) 1.880 (12.8%) 975 (6.7%) 9.505 (64.9%) 7.460 (51.0%) 4.856 (33.2%) 2.757 (18.8%) 1.568 (10.7%) 11.563 (79.0%) 213 (1.5%) 5.334 (36.4%) 8.676 (59.3%) 5.554 (38.0%) 309 (21%) 5.125 (35.0%) 1.838 (12.6%) 384 (2.6%) 1.995 (13.6%) 620 (4.2%) 1.2348 (84.4%) 2.412 (16.5%) | 0.0% (-0.1%, 0.1%) 0.1% (-0.0%, 0.3%) -0.12 (-0.14, -0.11) -(-,-) -(-,- | 34 (0.3%) 89 (0.7%) 229 (0.89) 2.00 [2.00, 3.00] 1.00, 6.00 6.341 (51.4%) 4.156 (33.7%) 3.182 (25.8%) 1.408 (11.4%) 862 (7.0%) 8.183 (66.3%) 5.415 (43.9%) 4.447 (36.0%) 2.061 (16.7%) 1.381 (11.2%) 9.764 (79.1%) 154 (1.2%) 4.481 (36.3%) 7.143 (57.9%) 4.722 (38.3%) 244 (20%) 4.140 (33.6%) 1.458 (11.8%) 312 (2.5%) 1.612 (13.1%) 540 (4.4%) 10.340 (83.8%) 1,931 (15.6%) | 29 (0.2%) 89 (0.7%) 228 (0.89) 2.00 [2.00, 3.00] 1.00, 6.00 6.364 (51.6%) 4,126 (33.4%) 3,097 (25.1%) 1.361 (11.0%) 825 (6.7%) 8.174 (66.2%) 5,377 (43.6%) 4,337 (35.1%) 2,018 (16.4%) 1,303 (10.6%) 9,678 (78.4%) 177 (1.4%) 4,473 (36.3%) 7,755 (38.1%) 262 (21%) 4,101 (33.2%) 1,437 (11.6%) 311 (2.5%) 1,605 (13.0%) 525 (4.3%) 1,031 (83.6%) 1,910 (15.5%) | 0.0% (-0.1%, 0.2%) 0.0% (-0.1%, 0.2%) 0.0% (-0.2%, 0.2%) 0.01 (-0.01, 0.04) -(-, -) -( |
| Bowel obstruction; n (%) Gastroparesis; n (%) Number of antidiabetic drugs on CEDmean (sd)median (IQR)min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of SGLT-2; n (%) Concomitant use or initiation of SGLT-2; n (%) Concomitant use or initiation of SGLT-2; n (%) Past use of Metformin; n (%) Past use of Insulins; n (%) Past use of Insulins; n (%) Past use of Sulfonylureas; n (%) Past use of Sulfonylureas; n (%) Past use of Any other glucose-lowering drugs; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ARNI; n (%) Thiazides; n (%) Beta-blockers; n (%) Calcium channel blockers; n (%) Digoxin / Digitoxin; n (%) Loop diuretics; n (%) Other diuretics; n (%) Nitrates; n (%) Nitrates; n (%) Anti-arrhythmics; n (%) Statins; n (%) Antiplatelet medications; n (%) Antiplatelet medications; n (%) Antiplatelet medications; n (%) | 167 (0.3%) 533 (0.8%) 219 (0.83) 200 [2.00, 3.00] 1.00, 6.00 36,599 (57.9%) 10,558 (16.7%) 20,522 (32.5%) 3,585 (5.7%) 41,72 (6.6%) 42,319 (67.0%) 14,679 (23.2%) 6,211 (9.8%) 49,068 (77.7%) 678 (11%) 22,378 (35.4%) 36,685 (58.1%) 25,814 (40.9%) 1,667 (26.%) 20,432 (32.3%) 6,557 (10.4%) 1,769 (2.8%) 7,852 (12.4%) 2,921 (4.6%) 51,100 (80.9%) 8,635 (13.7%) 10,621 (16.8%) | 36 (0.2%) 107 (0.7%) 107 (0.7%) 2.32 (0.90) 2.00 (2.00, 3.00) 1.00, 6.00 7.195 (49.2%) 5.854 (40.0%) 3.386 (23.1%) 1.880 (12.8%) 9.505 (64.9%) 7.460 (51.0%) 4.856 (33.2%) 2.757 (18.8%) 1.568 (10.7%) 11.563 (79.9%) 213 (1.5%) 5.334 (36.4%) 8.676 (59.3%) 5.554 (38.0%) 3.90 (2.1%) 5.125 (35.0%) 1.838 (12.6%) 3.84 (2.6%) 1.995 (13.6%) 620 (4.2%) 1.2,18.6%) 620 (4.2%) 1.2,18.6%) 620 (4.2%) 1.2,18.6%) 620 (4.2%) 1.2,18.6%) 620 (4.2%) | 0.0% (-0.1%, 0.1%) 0.1% (-0.0%, 0.3%) 0.12 (-0.14, -0.11) -(.,-) | 34 (0.3%) 89 (0.7%) 229 (0.89) 200 (2.00, 3.00) 1.00, 6.00 6.341 (51.4%) 4.156 (33.7%) 3.182 (25.8%) 1.408 (11.4%) 862 (7.0%) 8.183 (66.3%) 5.415 (43.9%) 4.447 (36.0%) 2.061 (16.7%) 1.381 (11.2%) 9,764 (79.1%) 154 (12.9%) 4.481 (36.3%) 7.143 (57.9%) 4,722 (38.3%) 1,472 (38.3%) 1,458 (11.8%) 312 (2.5%) 1,138 (11.9%) 1,145 (11.9%) 1,140 (33.6%) 1,145 (11.9%) 1,141 (11.1%) | 29 (0.2%) 89 (0.7%) 228 (0.89) 2.00 (2.00, 3.00) 1.00, 6.00 6.364 (61.6%) 4,126 (33.4%) 3,0.97 (25.1%) 1,361 (11.0%) 825 (6.7%) 8,174 (66.2%) 5,377 (43.6%) 4,337 (35.1%) 2,018 (16.4%) 1,303 (10.6%) 9,678 (78.4%) 177 (1.4%) 4,473 (36.3%) 4,705 (38.1%) 262 (2.1%) 4,101 (33.2%) 1,437 (11.6%) 311 (2.5%) 1,605 (13.0%) 525 (4.3%) 10,319 (83.6%) 1,910 (15.5%) 2,094 (17.0%) | 0.0% (-0.1%, 0.2%) 0.0% (-0.1%, 0.2%) 0.0% (-0.2%, 0.2%) 0.01 (-0.01, 0.04) -(·, ·) -( |
| Bowel obstruction; n (%) Gastroparesis; n (%) Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Past use of Metformin; n (%) Past use of Insulins; n (%) Past use of Insulins; n (%) Past use of Insulins; n (%) Past use of Sulfonylureas; n (%) Past use of Sulfonylureas; n (%) Past use of Any other glucose-lowering drugs; n (%) Past use of Any other glucose-lowering drugs; n (%) Past use of Any other glucose-lowering drugs; n (%) Calcium channel blockers; n (%) Digoxin / Digitoxin; n (%) Loop diuretics; n (%) Unop diuretics; n (%) Intravenous diuretics; n (%) Intravenous diuretics; n (%) Nitrates; n (%) Anti-arrhythmics; n (%) Statins; n (%) PCSK9 inhibitors and other lipid-lowering drugs; n (%) Oral anticoagulants; n (%) Oral anticoagulants; n (%) | 167 (0.3%) 533 (0.8%) 219 (0.83) 2.00 [2.00, 3.00] 1.00, 6.00 36,599 (57.9%) 10,558 (16.7%) 20,522 (32.5%) 3.585 (5.7%) 41,72 (6.6%) 42,319 (67.0%) 14,679 (23.2%) 26,424 (41.8%) 5,619 (8.9%) 6,211 (9.8%) 49,068 (77.7%) 678 (11%) 22,378 (35.4%) 36,685 (58.1%) 25,814 (40.9%) 1,667 (2.6%) 20,642 (32.3%) 6,557 (10.4%) 1,769 (2.8%) 7,852 (12.4%) 2,921 (4.6%) 51,100 (80.9%) 8,635 (13.7%) 10,621 (16.8%) 11,779 (18.6%) | 36 (0.2%) 107 (0.7%) 107 (0.7%) 2.32 (0.90) 2.00 [2.00, 3.00] 1.00, 6.00 7.195 (49.2%) 5.854 (40.0%) 3.386 (23.1%) 1.880 (12.8%) 9.505 (64.9%) 7.460 (51.0%) 4.856 (33.2%) 2.757 (18.8%) 1.568 (10.7%) 11,563 (79.0%) 2.13 (1.5%) 5.334 (36.4%) 8.676 (59.3%) 5.554 (38.0%) 3.90 (2.1%) 5,125 (35.0%) 1.838 (12.6%) 384 (2.6%) 1.838 (12.6%) 384 (2.6%) 1.995 (13.6%) 620 (4.2%) 12.342 (16.5%) 2.412 (16.5%) 2.571 (17.6%) 2.721 (18.6%) | 0.0% (-0.1%, 0.1%) 0.1% (-0.0%, 0.3%) 0.12 (-0.14, -0.11) -(.,-) | 34 (0.3%) 89 (0.7%) 229 (0.89) 200 (2.00, 3.00) 1.00, 6.00 6.341 (51.4%) 4.156 (33.7%) 3.182 (25.8%) 1,408 (11.4%) 862 (7.0%) 8.183 (66.3%) 5.415 (43.9%) 4.447 (36.0%) 2.061 (16.7%) 1,381 (11.2%) 9,764 (79.1%) 154 (12.%) 4,481 (36.3%) 7,143 (57.9%) 4,722 (38.3%) 244 (2.0%) 4,140 (33.6%) 1,458 (11.8%) 312 (25.9%) 1,612 (13.1%) 540 (4.4%) 10,340 (83.8%) 1,931 (15.6%) 2,114 (17.1%) 2,281 (18.5%) | 29 (0.2%) 89 (0.7%) 228 (0.89) 2.00 (2.00, 3.00) 1.00, 6.00 6.364 (51.6%) 4,126 (33.4%) 3,0.97 (25.1%) 1,361 (11.0%) 825 (6.7%) 8,174 (66.2%) 5,377 (43.6%) 4,337 (35.1%) 2,018 (16.4%) 1,303 (10.6%) 9,678 (78.4%) 1,77 (14.%) 4,473 (36.3%) 7,158 (58.0%) 4,705 (38.1%) 262 (2.1%) 4,101 (33.2%) 1,437 (11.6%) 311 (2.5%) 1,605 (13.0%) 525 (4.3%) 10,319 (83.6%) 1,910 (15.5%) 2,094 (17.0%) 2,270 (18.4%) | 0.0% (-0.1%, 0.2%) 0.0% (-0.1%, 0.2%) 0.0% (-0.2%, 0.2%) 0.01 (-0.01, 0.04) -(·,·) -(· |
| Bowel obstruction; n (%) Gastroparesis; n (%) Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of SGLT-2i; n (%) Concomitant use or initiation of SGLT-2i; n (%) Concomitant use or initiation of SGLT-2i; n (%) Past use of Metformin; n (%) Past use of Insulins; n (%) Past use of Insulins; n (%) Past use of Sulfonylureas; n (%) Past use of Sulfonylureas; n (%) Past use of Any other glucose-lowering drugs; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ARNI; n (%) Thiazides; n (%) Beta-blockers; n (%) Digoxin / Digitoxin; n (%) Digoxin / Digitoxin; n (%) Loop diuretics; n (%) Other diuretics; n (%) Nitrates; n (%) Nitrates; n (%) Anti-arrhythmics; n (%) Statins; n (%) Anti-arrhythmics; n (%) Antiplatelet medications; n (%) Antiplatelet medications; n (%) Antiplatelet medications; n (%) | 167 (0.3%) 533 (0.8%) 219 (0.83) 200 [2.00, 3.00] 1.00, 6.00 36,599 (57.9%) 10,558 (16.7%) 20,522 (32.5%) 3,585 (5.7%) 41,72 (6.6%) 42,319 (67.0%) 14,679 (23.2%) 6,211 (9.8%) 49,068 (77.7%) 678 (11%) 22,378 (35.4%) 36,685 (58.1%) 25,814 (40.9%) 1,667 (26.%) 20,432 (32.3%) 6,557 (10.4%) 1,769 (2.8%) 7,852 (12.4%) 2,921 (4.6%) 51,100 (80.9%) 8,635 (13.7%) 10,621 (16.8%) | 36 (0.2%) 107 (0.7%) 107 (0.7%) 2.32 (0.90) 2.00 (2.00, 3.00) 1.00, 6.00 7.195 (49.2%) 5.854 (40.0%) 3.386 (23.1%) 1.880 (12.8%) 9.505 (64.9%) 7.460 (51.0%) 4.856 (33.2%) 2.757 (18.8%) 1.568 (10.7%) 11.563 (79.9%) 213 (1.5%) 5.334 (36.4%) 8.676 (59.3%) 5.554 (38.0%) 3.90 (2.1%) 5.125 (35.0%) 1.838 (12.6%) 3.84 (2.6%) 1.995 (13.6%) 620 (4.2%) 1.2,18.6%) 620 (4.2%) 1.2,18.6%) 620 (4.2%) 1.2,18.6%) 620 (4.2%) 1.2,18.6%) 620 (4.2%) | 0.0% (-0.1%, 0.1%) 0.1% (-0.0%, 0.3%) 0.12 (-0.14, -0.11) -(.,-) | 34 (0.3%) 89 (0.7%) 229 (0.89) 200 (2.00, 3.00) 1.00, 6.00 6.341 (51.4%) 4.156 (33.7%) 3.182 (25.8%) 1.408 (11.4%) 862 (7.0%) 8.183 (66.3%) 5.415 (43.9%) 4.447 (36.0%) 2.061 (16.7%) 1.381 (11.2%) 9,764 (79.1%) 154 (12.9%) 4.481 (36.3%) 7.143 (57.9%) 4,722 (38.3%) 1,472 (38.3%) 1,458 (11.8%) 312 (2.5%) 1,138 (11.9%) 1,145 (11.9%) 1,140 (33.6%) 1,145 (11.9%) 1,141 (11.1%) | 29 (0.2%) 89 (0.7%) 228 (0.89) 2.00 (2.00, 3.00) 1.00, 6.00 6.364 (61.6%) 4,126 (33.4%) 3,0.97 (25.1%) 1,361 (11.0%) 825 (6.7%) 8,174 (66.2%) 5,377 (43.6%) 4,337 (35.1%) 2,018 (16.4%) 1,303 (10.6%) 9,678 (78.4%) 177 (1.4%) 4,473 (36.3%) 4,705 (38.1%) 262 (2.1%) 4,101 (33.2%) 1,437 (11.6%) 311 (2.5%) 1,605 (13.0%) 525 (4.3%) 10,319 (83.6%) 1,910 (15.5%) 2,094 (17.0%) | 0.0% (-0.1%, 0.2%) 0.0% (-0.1%, 0.2%) 0.01 (-0.01, 0.04) -(·, ·) -(·, |

| | • | • | • | • | • | |
|---|---|---|---|---|---|---|
| Oral corticosteroids; n (%) | 14,565 (23.0%) | 3,552 (24.3%) | -1.2% (-2.0%, -0.4%) | 2,995 (24.3%) | 2,964 (24.0%) | 0.3% (-0.8%, 1.3%) |
| Osteoporosis agents (incl. bisphosphonates); n (%) | 2,766 (4.4%) | 501 (3.4%) | 1.0% (0.6%, 1.3%) | 456 (3.7%) | 446 (3.6%) | 0.1% (-0.4%, 0.6%) |
| Opioids; n (%) | 23,761 (37.6%) | 5,985 (40.9%) | -3.3% (-4.2%, -2.4%) | 4,980 (40.4%) | 4,939 (40.0%) | 0.3% (-0.9%, 1.6%) |
| Anti-depressants; n (%) | 23,093 (36.5%) | 6,226 (42.5%) | -6.0% (-6.9%, -5.1%) | 5,176 (41.9%) | 5,107 (41.4%) | 0.6% (-0.7%, 1.8%) |
| Antipsychotics; n (%) | 3,060 (4.8%) | 602 (4.1%) | 0.7% (0.4%, 1.1%) | 510 (4.1%) | 518 (4.2%) | -0.1% (-0.6%, 0.4%) |
| Anxiolytics/hypnotics, benzos; n (%) | 13,290 (21.0%) | 3,248 (22.2%) | -1.2% (-1.9%, -0.4%) | 2,782 (22.5%) | 2,713 (22.0%) | 0.6% (-0.5%, 1.6%) |
| Dementia medications; n (%) | 3,407 (5.4%) | 450 (3.1%) | 2.3% (2.0%, 2.7%) | 381 (3.1%) | 405 (3.3%) | -0.2% (-0.6%, 0.3%) |
| Urinary tract infections antibiotics; n (%) | 33,868 (53.6%) | 8,134 (55.6%) | -2.0% (-2.9%, -1.1%) | 6,873 (55.7%) | 6,804 (55.1%) | 0.6% (-0.7%, 1.8%) |
| Laxatives; n (%) | 3,633 (5.7%) | 614 (4.2%) | 1.6% (1.2%, 1.9%) | 535 (4.3%) | 518 (4.2%) | 0.1% (-0.4%, 0.7%) |
| Number of distinct medications | | | | | | |
| mean (sd) | 14.85 (6.86) | 16.28 (6.83) | -1.43 (-1.55, -1.31) | 15.96 (7.01) | 15.84 (6.71) | 0.11 (-0.06, 0.28) |
| median [IQR] | 14.00 [10.00, 19.00] | 15.00 [11.00, 20.00] | - (-, -) | 15.00 [11.00, 20.00] | 15.00 [11.00, 20.00] | - (-, -) |
| min. max | 1.00, 64.00 | 1.00. 56.00 | - (-, -) | 1.00, 64.00 | 1.00, 56.00 | - (-, -) |
| Number of office visits | | | ( ) / | | | (,,, |
| mean (sd) | 11.68 (8.17) | 13.48 (8.56) | -1.81 (-1.96, -1.66) | 13.00 (9.01) | 12.96 (8.16) | 0.04 (-0.18, 0.25) |
| median [IQR] | 10.00 [6.00, 16.00] | 12.00 [7.00, 18.00] | - (-, -) | 11.00 [7.00, 17.00] | 11.00 [7.00, 17.00] | - (-, -) |
| min, max | 0.00, 211.00 | 0.00.145.00 | - (-, -) | 0.00, 211.00 | 0.00.98.00 | - (-, -) |
| Number of endocrinologist visits | 0.00, 211.00 | 0.00,143.00 | (, ) | 0.00, 211.00 | 0.00, 30.00 | ( , / |
| | 0.40 (1.36) | 0.96 (1.99) | -0.56 (-0.59, -0.52) | 0.72 (2.08) | 0.75 (1.64) | -0.03 (-0.07, 0.02) |
| mean (sd) | 0.40 (1.36) | | | 0.72 (2.08) | | |
| median [IQR] | | 0.00 [0.00, 1.00] | - (-, -) | | 0.00 [0.00, 1.00] | - (-, -) |
| min, max | 0.00, 66.00 | 0.00, 45.00 | - (-, -) | 0.00, 64.00 | 0.00, 28.00 | - (-, -) |
| Number of cardiologist visits | 225 (4.00) | 217/274 | 0.10 (0.11, 0.05) | 0.15 (0.00) | 214 (2.75) | 0.01 / 0.00 0.10 |
| mean (sd) | 2.35 (4.00) | 2.17 (3.74) | 0.18 (0.11, 0.25) | 2.15 (3.63) | 2.14 (3.75) | 0.01 (-0.08, 0.10) |
| median [IQR] | 1.00 [0.00, 3.00] | 1.00 [0.00, 3.00] | - (-, -) | 1.00 [0.00, 3.00] | 1.00 [0.00, 3.00] | - (-, -) |
| min, max | 0.00, 102.00 | 0.00, 62.00 | - (-, -) | 0.00, 49.00 | 0.00, 62.00 | - (-, -) |
| Number of internal/family medicine visits | | | | | | |
| mean (sd) | 7.29 (8.08) | 6.48 (6.65) | 0.81 (0.69, 0.94) | 6.52 (6.87) | 6.52 (6.74) | -0.00 (-0.17, 0.17) |
| median [IQR] | 5.00 [2.00, 10.00] | 5.00 [2.00, 9.00] | - (-, -) | 5.00 [2.00, 9.00] | 5.00 [2.00, 9.00] | - (-, -) |
| min, max | 0.00, 142.00 | 0.00, 84.00 | - (-, -) | 0.00, 125.00 | 0.00, 84.00 | - (-, -) |
| Number of Electrocardiograms (ECG/EKG) | | | | | | |
| mean (sd) | 1.74 (2.46) | 1.53 (2.19) | 0.21 (0.17, 0.25) | 1.54 (2.13) | 1.53 (2.22) | 0.01 (-0.05, 0.06) |
| median [IQR] | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | - (-, -) | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | - (-, -) |
| min, max | 0.00, 87.00 | 0.00, 38.00 | - (-, -) | 0.00, 31.00 | 0.00, 38.00 | - (-, -) |
| Number of Echocardiograms | | | | | | |
| mean (sd) | 0.53 (0.92) | 0.49 (0.86) | 0.05 (0.03, 0.06) | 0.48 (0.88) | 0.48 (0.86) | -0.00 (-0.03, 0.02) |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | - (-, -) | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | - (-, -) |
| min, max | 0.00, 23.00 | 0.00, 16.00 | - (-, -) | 0.00, 21.00 | 0.00, 16.00 | - (-, -) |
| Out-of-pocket medication cost | | | | | | |
| mean (sd) | 677.14 (841.58) | 1,070.64 (1,052.97) | -393.50 (-411.78, -375.22) | 950.03 (1,059.80) | 949.95 (941.67) | 0.08 (-24.93, 25.10) |
| median [IQR] | 424.38 [97.40, 952.26] | 767.08 [221.78, 1,614.22] | - (-, -) | 698.52 [176.09, 1,372.64] | 682.14 [188.49, 1,376.07] | - (-, -) |
| min, max | 0.00, 38,700.40 | 0.00, 23,893.53 | - (-, -) | 0.00, 38,700.40 | 0.00, 10,288.88 | - (-, -) |
| Unique brand medicines | | | ( ) / | | | ( ) / |
| mean (sd) | 15.18 (7.13) | 16.68 (7.13) | -1.51 (-1.64, -1.38) | 16.34 (7.32) | 16.23 (7.02) | 0.11 (-0.07, 0.29) |
| median [IQR] | 14.00 [10.00, 19.00] | 16.00 [12.00, 21.00] | - (-, -) | 15.00 [11.00, 20.00] | 15.00 [11.00, 20.00] | - (-, -) |
| min, max | 1.00, 73.00 | 1.00, 60.00 | - (-, -) | 1.00, 73.00 | 1.00, 60.00 | - (-, -) |
| Unique generic medicines | 1.00, 73.00 | 1.00, 00.00 | - (-, -) | 1.00, 73.00 | 1.00, 00.00 | -(57 |
| mean (sd) | 14.85 (6.86) | 16.28 (6.83) | -1.43 (-1.55, -1.31) | 15.96 (7.01) | 15.84 (6.71) | 0.11 (-0.06, 0.28) |
| | 14.00 [10.00, 19.00] | 15.00 [11.00, 20.00] | - (-, -) | 15.00 [11.00, 20.00] | 15.00 [11.00, 20.00] | - (-, -) |
| median [IQR] | | | | | 15.00 [11.00, 20.00] | - (-, -) |
| · | | | ( ) / | | 100 5000 | ( ) |
| min, max | 1.00, 64.00 | 1.00, 56.00 | - (-, -) | 1.00, 64.00 | 1.00, 56.00 | - (-, -) |
| Colonoscopy Sigmoidoscopy; n (%) | 1.00, 64.00<br>6,380 (10.1%) | 1.00, 56.00<br>1,697 (11.6%) | - (-, -)<br>-1.5% (-2.1%, -0.9%) | 1.00, 64.00<br>1,376 (11.2%) | 1,368 (11.1%) | 0.1% (-0.7%, 0.9%) |
| Colonoscopy Sigmoidoscopy; n (%) Flu Pneumococcal vaccine; n (%) | 1.00, 64.00<br>6,380 (10.1%)<br>7,895 (12.5%) | 1.00, 56.00<br>1,697 (11.6%)<br>1,593 (10.9%) | - (-, -)<br>-1.5% (-2.1%, -0.9%)<br>1.6% (1.0%, 2.2%) | 1.00, 64.00<br>1,376 (11.2%)<br>1,376 (11.2%) | 1,368 (11.1%)<br>1,349 (10.9%) | 0.1% (-0.7%, 0.9%)<br>0.2% (-0.6%, 1.0%) |
| Colonoscopy Sigmoidoscopy; n (%) Flu Pneumococcal vaccine; n (%) Pap smear; n (%) | 1.00, 64.00<br>6,380 (10.1%)<br>7,895 (12.5%)<br>2,376 (3.8%) | 1.00, 56.00<br>1.697 (11.6%)<br>1.593 (10.9%)<br>700 (4.8%) | -(-, -)<br>-1.5% (-2.1%, -0.9%)<br>1.6% (1.0%, 2.2%)<br>-1.0% (-1.4%, -0.6%) | 1.00, 64.00<br>1,376 (11.2%)<br>1,376 (11.2%)<br>640 (5.2%) | 1,368 (11.1%)<br>1,349 (10.9%)<br>578 (4.7%) | 0.1% (-0.7%, 0.9%)<br>0.2% (-0.6%, 1.0%)<br>0.5% (-0.0%, 1.1%) |
| Colonoscopy Sigmoidoscopy; n (%) Flu Pneumococcal vaccine; n (%) Pap smear; n (%) PSA test; n (%) | 1.00, 64.00<br>6,380 (10.1%)<br>7,895 (12.5%)<br>2,376 (3.8%)<br>12,330 (19.5%) | 1.00, 56.00<br>1.697 (11.6%)<br>1.593 (10.9%)<br>700 (4.8%)<br>3,321 (22.7%) | -(-, -)<br>-1.5% (-2.1%, -0.9%)<br>1.6% (1.0%, 2.2%)<br>-1.0% (-1.4%, -0.6%)<br>-3.2% (-3.9%, -2.4%) | 1.00, 64.00<br>1,376 (11.2%)<br>1,376 (11.2%)<br>640 (5.2%)<br>2,692 (21.8%) | 1,368 (11.1%)<br>1,349 (10.9%)<br>578 (4.7%)<br>2,740 (22.2%) | 0.1% (-0.7%, 0.9%)<br>0.2% (-0.6%, 1.0%)<br>0.5% (-0.0%, 1.1%)<br>-0.4% (-1.4%, 0.7%) |
| Colonoscopy Sigmoidoscopy; n (%) Flu Pneumococcal vaccine; n (%) Pap smear; n (%) PSA test n (%) Fecal occult blood test; n (%) | 1.00, 64.00<br>6,380 (10.1%)<br>7,895 (12.5%)<br>2,376 (3.8%)<br>12,330 (19.5%)<br>4,720 (7.5%) | 1.00, 56.00<br>1.697 (11.6%)<br>1.593 (10.9%)<br>700 (4.8%)<br>3.321 (22.7%)<br>897 (6.1%) | -(-,-)<br>-1.5% (-2.1%, -0.9%)<br>1.6% (1.0%, 2.2%)<br>-1.0% (-1.4%, -0.6%)<br>-3.2% (-3.9%, -2.4%)<br>1.3% (0.9%, 1.8%) | 1.00, 64.00<br>1.376 (11.2%)<br>1.376 (11.2%)<br>640 (5.2%)<br>2.692 (21.8%)<br>788 (6.4%) | 1,368 (11.1%)<br>1,349 (10.9%)<br>578 (4.7%)<br>2,740 (22.2%)<br>789 (6.4%) | 0.1% (-0.7%, 0.9%)<br>0.2% (-0.6%, 1.0%)<br>0.5% (-0.0%, 1.1%)<br>-0.4% (-1.4%, 0.7%)<br>-0.0% (-0.6%, 0.6%) |
| Colonoscopy Sigmoidoscopy; n (%) Flu Pneumococcal vaccine; n (%) Pap smear; n (%) PSA test; n (%) Fecal occult blood test; n (%) Bone mineral density tests; n (%) | 1.00, 64.00<br>6,380 (10.1%)<br>7,895 (12.5%)<br>2,376 (3.8%)<br>12,330 (19.5%)<br>4,720 (7.5%)<br>5,240 (8.3%) | 1.00, 56.00<br>1.697 (11.6%)<br>1.593 (10.9%)<br>700 (4.8%)<br>3.321 (22.7%)<br>897 (6.1%)<br>1.397 (9.5%) | -(,-)<br>-1.5% (-2.1%, -0.9%)<br>1.6% (1.0%, 2.2%)<br>-1.0% (-1.4%, -0.6%)<br>-3.2% (-3.9%, -2.4%)<br>1.3% (0.9%, 1.8%)<br>-1.3% (-1.8%, -0.7%) | 1.00, 64.00<br>1,376 (11.2%)<br>1,376 (11.2%)<br>640 (5.2%)<br>2.692 (21.8%)<br>788 (6.4%)<br>1,169 (9.5%) | 1,368 (11.1%)<br>1,349 (10.9%)<br>578 (4.7%)<br>2,740 (22.2%)<br>789 (6.4%)<br>1,162 (9.4%) | 0.1% (-0.7%, 0.9%)<br>0.2% (-0.6%, 1.0%)<br>0.5% (-0.0%, 1.1%)<br>-0.4% (-1.4%, 0.7%)<br>-0.0% (-0.6%, 0.6%)<br>0.1% (-0.7%, 0.8%) |
| Colonoscopy Sigmoidoscopy; n (%) Flu Pneumococcal vaccine; n (%) Pap smear, n (%) PSA test; n (%) Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) | 1.00, 64.00<br>6.380 (10.1%)<br>7.895 (12.5%)<br>2.376 (3.8%)<br>12,330 (19.5%)<br>4.720 (7.5%)<br>5.240 (8.3%)<br>12,802 (20.3%) | 1.00, 56.00<br>1,697 (11.6%)<br>1.593 (10.9%)<br>700 (4.8%)<br>3.321 (22.7%)<br>897 (6.1%)<br>1.397 (9.5%)<br>3,463 (23.7%) | -(-,-)<br>-1.5% (-21%, -0.9%)<br>1.6% (1.0%, 2.2%)<br>-1.0% (-1.4%, -0.6%)<br>-3.2% (-3.9%, -2.4%)<br>1.3% (0.9%, 1.8%)<br>-1.3% (-1.8%, -0.7%)<br>-3.4% (-4.2%, -2.6%) | 1.00, 64.00<br>1,376 (11.2%)<br>1,376 (11.2%)<br>640 (5.2%)<br>2,692 (21.8%)<br>788 (6.4%)<br>1,169 (9.5%)<br>2,938 (23.8%) | 1,368 (11.1%)<br>1,349 (10.9%)<br>578 (4.7%)<br>2,740 (22.2%)<br>789 (6.4%)<br>1,162 (9.4%)<br>2,874 (23.3%) | 0.1% (-0.7%, 0.9%)<br>0.2% (-0.6%, 1.0%)<br>0.5% (-0.0%, 1.1%)<br>-0.4% (-1.4%, 0.7%)<br>-0.0% (-0.6%, 0.6%)<br>0.1% (-0.7%, 0.8%)<br>0.5% (-0.5%, 1.6%) |
| Colonoscopy Sigmoidoscopy; n (%) Flu Pneumococcal vaccine; n (%) Pap smear; n (%) PSA test; n (%) Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) | 1.00, 64.00<br>6,380 (10.1%)<br>7,895 (12.5%)<br>2,376 (3.8%)<br>12,330 (19.5%)<br>4,720 (7.5%)<br>5,240 (8.3%) | 1.00, 56.00<br>1.697 (11.6%)<br>1.593 (10.9%)<br>700 (4.8%)<br>3.321 (22.7%)<br>897 (6.1%)<br>1.397 (9.5%) | -(,-)<br>-1.5% (-2.1%, -0.9%)<br>1.6% (1.0%, 2.2%)<br>-1.0% (-1.4%, -0.6%)<br>-3.2% (-3.9%, -2.4%)<br>1.3% (0.9%, 1.8%)<br>-1.3% (-1.8%, -0.7%) | 1.00, 64.00<br>1,376 (11.2%)<br>1,376 (11.2%)<br>640 (5.2%)<br>2.692 (21.8%)<br>788 (6.4%)<br>1,169 (9.5%) | 1,368 (11.1%)<br>1,349 (10.9%)<br>578 (4.7%)<br>2,740 (22.2%)<br>789 (6.4%)<br>1,162 (9.4%) | 0.1% (-0.7%, 0.9%)<br>0.2% (-0.6%, 1.0%)<br>0.5% (-0.0%, 1.1%)<br>-0.4% (-1.4%, 0.7%)<br>-0.0% (-0.6%, 0.6%)<br>0.1% (-0.7%, 0.8%) |
| Colonoscopy Sigmoidoscopy; n (%) Flu Pneumococcal vaccine; n (%) Pap smear, n (%) PSA test; n (%) Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) | 1.00, 64.00<br>6.380 (10.1%)<br>7.895 (12.5%)<br>2.376 (3.8%)<br>12,330 (19.5%)<br>4,720 (7.5%)<br>5,240 (8.3%)<br>12,802 (20.3%)<br>4,273 (6.8%) | 1.00, 56.00<br>1.697 (11.6%)<br>1.593 (10.9%)<br>700 (4.8%)<br>3.321 (22.7%)<br>897 (6.1%)<br>1,397 (9.5%)<br>3,463 (23.7%)<br>2,322 (15.9%) | -(-,-)<br>-15% (-21%, -0.9%)<br>16% (1.0%, 2.2%)<br>-1.0% (-1.4%, -0.6%)<br>-3.2% (-3.9%, -2.4%)<br>1.3% (0.9%, 1.8%)<br>-1.3% (-1.8%, -0.7%)<br>-3.4% (-4.2%, -2.6%)<br>-9.1% (-9.7%, -8.5%) | 100, 64.00<br>1,376 (11.2%)<br>1,376 (11.2%)<br>640 (5.2%)<br>2,692 (21.8%)<br>788 (6.4%)<br>1,169 (9.5%)<br>2,938 (23.8%)<br>1,685 (13.7%) | 1,368 (11.1%)<br>1,349 (10.9%)<br>578 (4.7%)<br>2,740 (22.2%)<br>789 (6.4%)<br>1,162 (9.4%)<br>2,874 (23.3%)<br>1,716 (13.9%) | 0.1% (-0.7%, 0.9%) 0.2% (-0.6%, 1.0%) 0.5% (-0.6%, 1.0%) 0.5% (-0.0%, 1.1%) -0.4% (-1.4%, 0.7%) -0.0% (-0.6%, 0.6%) 0.1% (-0.7%, 0.8%) 0.5% (-0.5%, 1.6%) -0.3% (-1.1%, 0.6%) |
| Colonoscopy Sigmoidoscopy; n (%) Flu Pneumococcal vaccine; n (%) Pap smear; n (%) PSA test; n (%) Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) | 1.00, 64.00<br>6.380 (10.1%)<br>7.895 (12.5%)<br>2.376 (3.8%)<br>12.330 (19.5%)<br>4.720 (7.5%)<br>5.240 (8.3%)<br>12,802 (20.3%)<br>4,273 (6.8%) | 1.00, 56.00<br>1.697 (11.6%)<br>1.593 (10.9%)<br>700 (4.8%)<br>3.321 (22.7%)<br>897 (6.1%)<br>1.397 (9.5%)<br>3.463 (23.7%)<br>2.322 (15.9%) | -(-,-)<br>-1.5% (-21%, -0.9%)<br>1.6% (1.0%, 2.2%)<br>-1.0% (-1.4%, -0.6%)<br>-3.2% (-3.9%, -2.4%)<br>1.3% (0.9%, 1.8%)<br>-1.3% (-1.8%, -0.7%)<br>-3.4% (-4.2%, -2.6%) | 100, 64.00<br>1,376 (11.2%)<br>1,376 (11.2%)<br>640 (5.2%)<br>2,692 (21.8%)<br>788 (6.4%)<br>1,169 (9.5%)<br>2,938 (23.8%)<br>1,685 (13.7%) | 1,368 (11.1%)<br>1,349 (10.9%)<br>578 (4.7%)<br>2,740 (22.2%)<br>789 (6.4%)<br>1,162 (9.4%)<br>2,874 (23.3%) | 0.1% (-0.7%, 0.9%)<br>0.2% (-0.6%, 1.0%)<br>0.5% (-0.0%, 1.1%)<br>-0.4% (-1.4%, 0.7%)<br>-0.0% (-0.6%, 0.6%)<br>0.1% (-0.7%, 0.8%)<br>0.5% (-0.5%, 1.6%) |
| Colonoscopy Sigmoidoscopy; n (%) Flu Pneumococcal vaccine; n (%) Pap smear; n (%) PSA test n (%) Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbAIC tests | 1.00, 64.00<br>6.380 (10.1%)<br>7.895 (12.5%)<br>2.376 (3.8%)<br>12,330 (19.5%)<br>4.720 (7.5%)<br>5.240 (8.3%)<br>12,802 (20.3%)<br>4.273 (6.8%)<br>2.71 (2.84)<br>3.00 (2.00, 3.00) | 1.00, 56.00<br>1.697 (11.6%)<br>1.593 (10.9%)<br>700 (4.8%)<br>3.321 (22.7%)<br>897 (6.1%)<br>1.397 (9.5%)<br>3.463 (23.7%)<br>2.322 (15.9%)<br>2.96 (2.04)<br>3.00 (2.00, 4.00) | -(-,-)<br>-1.5% (-2.1%, -0.9%)<br>1.6% (1.0%, 2.2%)<br>-1.0% (-1.4%, -0.6%)<br>-3.2% (-3.9%, -2.4%)<br>1.3% (0.9%, 1.8%)<br>-1.3% (-1.8%, -0.7%)<br>-3.4% (-4.2%, -2.6%)<br>-9.1% (-9.7%, -8.5%)<br>-0.25 (-0.29, -0.21)<br>-(-,-) | 1.00, 64.00<br>1,376 (11.2%)<br>1.376 (11.2%)<br>640 (5.2%)<br>2.692 (21.8%)<br>788 (6.4%)<br>1.169 (9.5%)<br>2.938 (23.8%)<br>1.685 (13.7%)<br>2.90 (3.32)<br>3.00 (2.00, 4.00) | 1,368 (11.1%) 1,349 (10.9%) 578 (4.7%) 2,740 (22.2%) 789 (6.4%) 1,162 (9.4%) 1,716 (13.9%) 2,89 (1.93) 3,00 (2.00, 4.00) | 0.1% (-0.7%, 0.9%) 0.2% (-0.6%, 1.0%) 0.5% (-0.0%, 1.1%) -0.4% (-1.4%, 0.7%) -0.0% (-0.6%, 0.6%) 0.1% (-0.7%, 0.8%) 0.5% (-0.5%, 1.6%) -0.3% (-1.1%, 0.6%) 0.01 (-0.06, 0.07) - (-, -) |
| Colonoscopy Sigmoidoscopy; n (%) Flu Pneumococcal vaccine; n (%) Pap smear; n (%) PSA test; n (%) Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbAIC testsmean (sd) | 1.00, 64.00<br>6.380 (10.1%)<br>7.895 (12.5%)<br>2.376 (3.8%)<br>12.330 (19.5%)<br>4.720 (7.5%)<br>5.240 (8.3%)<br>12,802 (20.3%)<br>4,273 (6.8%) | 1.00, 56.00<br>1.697 (11.6%)<br>1.593 (10.9%)<br>700 (4.8%)<br>3.321 (22.7%)<br>897 (6.1%)<br>1.397 (9.5%)<br>3.463 (23.7%)<br>2.322 (15.9%) | -(,-)<br>-1.5% (-2.1%, -0.9%)<br>1.6% (1.0%, 2.2%)<br>-1.0% (-1.4%, -0.6%)<br>-3.2% (-3.9%, -2.4%)<br>1.3% (0.9%, 1.8%)<br>-1.3% (-1.8%, -0.7%)<br>-3.4% (-4.2%, -2.6%)<br>-9.1% (-9.7%, -8.5%)<br>-0.25 (-0.29, -0.21) | 100, 64.00<br>1,376 (11.2%)<br>1,376 (11.2%)<br>640 (5.2%)<br>2,692 (21.8%)<br>788 (6.4%)<br>1,169 (9.5%)<br>2,938 (23.8%)<br>1,685 (13.7%) | 1,368 (11.1%)<br>1,349 (10.9%)<br>578 (4.7%)<br>2,740 (22.2%)<br>789 (6.4%)<br>1,162 (9.4%)<br>2,874 (23.3%)<br>1,716 (13.9%)<br>2,89 (1.93) | 0.1% (-0.7%, 0.9%)<br>0.2% (-0.6%, 1.0%)<br>0.5% (-0.0%, 1.1%)<br>0.5% (-0.0%, 1.1%)<br>-0.4% (-1.4%, 0.7%)<br>-0.0% (-0.6%, 0.6%)<br>0.1% (-0.7%, 0.8%)<br>0.5% (-0.5%, 1.6%)<br>-0.3% (-1.1%, 0.6%) |
| Colonoscopy Sigmoidoscopy; n (%) Flu Pneumococcal vaccine; n (%) Pap smear; n (%) PSA test; n (%) Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbA1C testsmean (sd)median [IQR] | 1.00, 64.00<br>6.380 (10.1%)<br>7.895 (12.5%)<br>2.376 (3.8%)<br>12,330 (19.5%)<br>4.720 (7.5%)<br>5.240 (8.3%)<br>12,802 (20.3%)<br>4.273 (6.8%)<br>2.71 (2.84)<br>3.00 (2.00, 3.00) | 1.00, 56.00<br>1.697 (11.6%)<br>1.593 (10.9%)<br>700 (4.8%)<br>3.321 (22.7%)<br>897 (6.1%)<br>1.397 (9.5%)<br>3.463 (23.7%)<br>2.322 (15.9%)<br>2.96 (2.04)<br>3.00 (2.00, 4.00) | -(-,-)<br>-1.5% (-2.1%, -0.9%)<br>1.6% (1.0%, 2.2%)<br>-1.0% (-1.4%, -0.6%)<br>-3.2% (-3.9%, -2.4%)<br>1.3% (0.9%, 1.8%)<br>-1.3% (-1.8%, -0.7%)<br>-3.4% (-4.2%, -2.6%)<br>-9.1% (-9.7%, -8.5%)<br>-0.25 (-0.29, -0.21)<br>-(-,-) | 1.00, 64.00<br>1,376 (11.2%)<br>1.376 (11.2%)<br>640 (5.2%)<br>2.692 (21.8%)<br>788 (6.4%)<br>1.169 (9.5%)<br>2.938 (23.8%)<br>1.685 (13.7%)<br>2.90 (3.32)<br>3.00 (2.00, 4.00) | 1,368 (11.1%) 1,349 (10.9%) 578 (4.7%) 2,740 (22.2%) 789 (6.4%) 1,162 (9.4%) 1,716 (13.9%) 2,89 (1.93) 3,00 (2.00, 4.00) | 0.1% (-0.7%, 0.9%) 0.2% (-0.6%, 1.0%) 0.5% (-0.0%, 1.1%) -0.4% (-1.4%, 0.7%) -0.0% (-0.6%, 0.6%) 0.1% (-0.7%, 0.8%) 0.5% (-0.5%, 1.6%) -0.3% (-1.1%, 0.6%) 0.01 (-0.06, 0.07) - (-, -) |
| Colonoscopy Sigmoidoscopy; n (%) Flu Pneumococcal vaccine; n (%) Pap smear; n (%) PSA test; n (%) Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbAIC testsmean (sd)median [UQR]min, max | 1.00, 64.00<br>6.380 (10.1%)<br>7.895 (12.5%)<br>2.376 (3.8%)<br>12,330 (19.5%)<br>4.720 (7.5%)<br>5.240 (8.3%)<br>12,802 (20.3%)<br>4.273 (6.8%)<br>2.71 (2.84)<br>3.00 (2.00, 3.00) | 1.00, 56.00<br>1.697 (11.6%)<br>1.593 (10.9%)<br>700 (4.8%)<br>3.321 (22.7%)<br>897 (6.1%)<br>1.397 (9.5%)<br>3.463 (23.7%)<br>2.322 (15.9%)<br>2.96 (2.04)<br>3.00 (2.00, 4.00) | -(-,-)<br>-1.5% (-2.1%, -0.9%)<br>1.6% (1.0%, 2.2%)<br>-1.0% (-1.4%, -0.6%)<br>-3.2% (-3.9%, -2.4%)<br>1.3% (0.9%, 1.8%)<br>-1.3% (-1.8%, -0.7%)<br>-3.4% (-4.2%, -2.6%)<br>-9.1% (-9.7%, -8.5%)<br>-0.25 (-0.29, -0.21)<br>-(-,-) | 1.00, 64.00<br>1,376 (11.2%)<br>1.376 (11.2%)<br>640 (5.2%)<br>2.692 (21.8%)<br>788 (6.4%)<br>1.169 (9.5%)<br>2.938 (23.8%)<br>1.685 (13.7%)<br>2.90 (3.32)<br>3.00 (2.00, 4.00) | 1,368 (11.1%) 1,349 (10.9%) 578 (4.7%) 2,740 (22.2%) 789 (6.4%) 1,162 (9.4%) 1,716 (13.9%) 2,89 (1.93) 3,00 (2.00, 4.00) | 0.1% (-0.7%, 0.9%) 0.2% (-0.6%, 1.0%) 0.5% (-0.0%, 1.1%) -0.4% (-1.4%, 0.7%) -0.0% (-0.6%, 0.6%) 0.1% (-0.7%, 0.8%) 0.5% (-0.5%, 1.6%) -0.3% (-1.1%, 0.6%) 0.01 (-0.06, 0.07) - (-, -) |
| Colonoscopy Sigmoidoscopy; n (%) Flu Pneumococcal vaccine; n (%) Pap smear; n (%) PSA test n (%) Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbAIC testsmean (sd)median [UR]min, max Lipid panels | 1.00, 64.00<br>6.380 (10.1%)<br>7.895 (12.5%)<br>2.376 (3.8%)<br>12,330 (19.5%)<br>4.720 (7.5%)<br>5.240 (8.3%)<br>12,802 (20.3%)<br>4,273 (6.8%)<br>2.71 (2.84)<br>3.00 [2.00, 3.00]<br>0.00, 215.00 | 1.00, 56.00<br>1.697 (11.6%)<br>1.593 (10.9%)<br>700 (4.8%)<br>3.321 (22.7%)<br>897 (6.1%)<br>1.397 (9.5%)<br>3.463 (23.7%)<br>2.322 (15.9%)<br>2.96 (2.04)<br>3.00 [2.00, 4.00]<br>0.00, 74.00 | -(-,-)<br>-15% (-21%, -0.9%)<br>1.6% (1.0%, 2.2%)<br>1.0% (-1.4%, -0.6%)<br>3.2% (-3.9%, -2.4%)<br>1.3% (0.9%, 1.8%)<br>-1.3% (-1.8%, -0.7%)<br>-3.4% (-4.2%, -2.6%)<br>-9.1% (-9.7%, -8.5%)<br>-0.25 (-0.29, -0.21)<br>-(-,-) | 1.00, 64.00<br>1.376 (11.2%)<br>640 (5.2%)<br>2.692 (21.8%)<br>788 (6.4%)<br>1.169 (9.5%)<br>2.938 (23.8%)<br>1.685 (13.7%)<br>2.90 (3.32)<br>3.00 (2.00, 4.00)<br>0.00, 163.00 | 1,368 (11.1%) 1,349 (10.9%) 578 (4.7%) 2,740 (22.2%) 789 (6.4%) 1,162 (9.4%) 2,874 (23.3%) 1,716 (13.9%) 2,89 (1.93) 3,00 [2.00, 4.00] 0,00, 74.00 | 0.1% (-0.7%, 0.9%) 0.2% (-0.6%, 1.0%) 0.5% (-0.0%, 1.1%) 0.5% (-0.0%, 1.1%) -0.4% (-1.4%, 0.7%) -0.0% (-0.6%, 0.6%) 0.1% (-0.7%, 0.8%) 0.5% (-0.5%, 1.6%) -0.3% (-1.1%, 0.6%) 0.11 (-0.06, 0.07) -(-, -) |
| Colonoscopy Sigmoidoscopy; n (%) Flu Pneumococcal vaccine; n (%) Pap smear, n (%) PSA test; n (%) PSA test; n (%) Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbAIC testsmean (sd)median [IQR]min, max Lipid panelsmean (sd) | 1.00, 64.00<br>6.380 (10.1%)<br>7.895 (12.5%)<br>2.376 (3.8%)<br>12.330 (19.5%)<br>4.720 (7.5%)<br>5.240 (8.3%)<br>12.802 (20.3%)<br>4.273 (6.8%)<br>2.71 (2.84)<br>3.00 [2.00, 3.00]<br>0.00, 215.00 | 1.00, 56.00<br>1.697 (11.6%)<br>1.593 (10.9%)<br>700 (4.8%)<br>3.321 (22.7%)<br>897 (6.1%)<br>1.397 (9.5%)<br>3.463 (23.7%)<br>2.322 (15.9%)<br>2.96 (2.04)<br>3.00 [2.00, 4.00]<br>0.00, 74.00 | -(-,-) -(5,-) -(1.9% (-2.1%, -0.9%) -(1.0% (-2.1%, -0.9%) -(1.0% (-1.4%, -0.6%) -(3.2% (-3.9%, -2.4%) -(3.3% (-1.8%, -0.7%) -(3.4% (-4.2%, -2.6%) -(9.1% (-9.7%, -8.5%) -(0.25 (-0.29, -0.21) -(-,-) -(-,-) -(1.0 (-0.14, -0.07) | 1.00, 64.00<br>1,376 (11.2%)<br>640 (5.2%)<br>640 (5.2%)<br>2692 (21.8%)<br>788 (6.4%)<br>1,169 (9.5%)<br>2,938 (23.8%)<br>1,685 (13.7%)<br>2.90 (3.32)<br>3.00 (2.00, 4.00)<br>0.00, 163.00 | 1,368 (11.1%) 1,349 (10.9%) 578 (4.7%) 2,740 (22.2%) 789 (6.4%) 1,162 (9.4%) 2,874 (23.3%) 1,716 (13.9%) 2,89 (1.93) 3.00 (2.00, 4.00) 0.00, 74.00 | 0.1% (-0.7%, 0.9%) 0.2% (-0.6%, 1.0%) 0.5% (-0.0%, 1.1%) 0.5% (-0.0%, 1.1%) 0.0% (-0.6%, 0.6%) 0.1% (-0.7%, 0.8%) 0.1% (-0.7%, 0.8%) 0.5% (-0.5%, 1.6%) 0.3% (-1.1%, 0.6%) 0.01 (-0.06, 0.07) -(-, -) -(-, -) 0.02 (-0.04, 0.07) |
| Colonoscopy Sigmoidoscopy; n (%) Flu Pneumococcal vaccine; n (%) Pap smear; n (%) PSA test; n (%) Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbALC testsmean (sd)median [IQR]min, max Lipid panelsmean (sd)median [IQR] | 1.00, 64.00<br>6.380 (10.1%)<br>7.895 (12.5%)<br>2.376 (3.8%)<br>12,330 (19.5%)<br>4.720 (7.5%)<br>5.240 (8.3%)<br>12,802 (20.3%)<br>4.273 (6.8%)<br>2.71 (2.84)<br>3.00 (2.00, 3.00)<br>0.00, 215.00<br>1.82 (2.15)<br>2.00 (1.00, 2.00) | 1.00, 56.00<br>1.697 (11.6%)<br>1.593 (10.9%)<br>700 (4.8%)<br>3.321 (22.7%)<br>897 (6.1%)<br>1.397 (9.5%)<br>3.463 (23.7%)<br>2.322 (15.9%)<br>2.96 (2.04)<br>3.00 (2.00, 4.00)<br>0.00, 74.00<br>1.92 (1.74)<br>2.00 (1.00, 3.00) | -(-,-) -(5% (-21% -0.9%) -(1.6% (1.0%, 2.2%) -(1.0% (1.4%, -0.6%) -(3.2% (-3.9%, -2.4%) -(3.9%, 1.8%) -(3.4% (-4.2%, -2.6%) -(3.4% (-4.2% (-4.2%) -(3.4% (-4.2% (-4.2%) -(3.4% (-4.2%) -(3.4% (-4.2% (-4.2%) -(3.4% (-4.2%) -(3 | 1.00, 64.00<br>1,376 (11.2%)<br>640 (5.2%)<br>2.692 (21.8%)<br>788 (6.4%)<br>1,169 (9.5%)<br>2,938 (23.8%)<br>1,685 (13.7%)<br>290 (3.32)<br>3.00 (2.00, 4.00)<br>0.00, 163.00<br>1.93 (2.68)<br>2.00 (1.00, 3.00) | 1,368 (111%) 1,349 (10.9%) 578 (4.7%) 2,740 (22.2%) 789 (6.4%) 1,162 (9.4%) 1,176 (13.9%) 2,874 (23.3%) 1,716 (13.9%) 2,89 (1.93) 3.00 (2.00, 4.00) 0.00, 74.00 1.91 (1.78) 2.00 (1.00, 3.00) | 0.1% (-0.7%, 0.9%) 0.2% (-0.6%, 1.0%) 0.5% (-0.0%, 1.1%) 0.5% (-0.0%, 1.1%) -0.4% (-1.4%, 0.7%) -0.0% (-0.6%, 0.6%) 0.1% (-0.7%, 0.8%) 0.5% (-0.5%, 1.6%) -0.3% (-1.1%, 0.6%) 0.01 (-0.06, 0.07) -(-, -) -(-, -) 0.02 (-0.04, 0.07) -(-, -) |

| mean (sd) | 0.11 (0.78) | 0.10 (0.53) | 0.01 (0.00, 0.03) | 0.09 (0.49) | 0.09 (0.51) | -0.00 (-0.01, 0.01) |
|---|---|---|---|---|---|---|
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) |
| min, max | 0.00, 59.00 | 0.00,16.00 | - (-, -) | 0.00, 16.00 | 0.00, 16.00 | - (-, -) |
| Natriuretic peptide tests | | | ( ) / | | | ( ) / |
| mean (sd) | 0.40 (1.88) | 0.38 (1.64) | 0.02 (-0.01, 0.05) | 0.38 (1.72) | 0.37 (1.63) | 0.01 (-0.04, 0.05) |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) |
| min, max | 0.00.193.00 | 0.00, 84.00 | - (-, -) | 0.00, 82.00 | 0.00, 84,00 | - (-, -) |
| Urine tests | | | | | | |
| mean (sd) | 1.73 (3.30) | 1.60 (2.82) | 0.13 (0.08, 0.18) | 1.61 (2.82) | 1.61 (2.91) | 0.00 (-0.07, 0.08) |
| median [IQR] | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | - (-, -) | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | - (-, -) |
| min, max | 0.00, 237.00 | 0.00, 98.00 | - (-, -) | 0.00, 105.00 | 0.00, 98.00 | - (-, -) |
| Combined comorbidity score | | | | | | |
| mean (sd) | 2.88 (2.95) | 2.66 (2.58) | 0.22 (0.17, 0.27) | 2.62 (2.60) | 2.62 (2.61) | -0.01 (-0.07, 0.06) |
| median [IQR] | 2.00 [1.00, 5.00] | 2.00 [1.00, 4.00] | - (-, -) | 2.00 [1.00, 4.00] | 2.00 [1.00, 4.00] | - (-, -) |
| min, max | -2.00, 17.00 | -2.00, 16.00 | - (-, -) | -2.00, 16.00 | -2.00, 16.00 | - (-, -) |
| Frailty Score | | | | | | |
| mean (sd) | 0.22 (0.08) | 0.22 (0.07) | 0.01 (0.01, 0.01) | 0.22 (0.07) | 0.22 (0.07) | -0.00 (-0.00, 0.00) |
| median [IQR] | 0.21 [0.17, 0.26] | 0.20 [0.17, 0.25] | - (-, -) | 0.20 [0.16, 0.25] | 0.20 [0.17, 0.25] | - (-, -) |
| min, max | 0.06, 0.69 | 0.07, 0.63 | - (-, -) | 0.06, 0.65 | 0.07, 0.63 | - (-, -) |
| Number of Hospitalizations | | | | | | |
| mean (sd) | 0.61 (1.19) | 0.41 (0.89) | 0.20 (0.18, 0.22) | 0.43 (0.91) | 0.43 (0.92) | 0.00 (-0.02, 0.03) |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | - (-, -) | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | - (-, -) |
| min, max | 0.00, 31.00 | 0.00, 12.00 | - (-, -) | 0.00, 11.00 | 0.00, 12.00 | - (-, -) |
| Any hospitalization within prior 91 days; n (%) | 9,448 (15.0%) | 1,147 (7.8%) | 7.1% (6.6%, 7.6%) | 1,072 (8.7%) | 1,061 (8.6%) | 0.1% (-0.6%, 0.8%) |
| Any hospitalization within prior 92-365 days; n (%) | 15,731 (24.9%) | 3,167 (21.6%) | 3.3% (2.5%, 4.0%) | 2,691 (21.8%) | 2,667 (21.6%) | 0.2% (-0.8%, 1.2%) |
| Number of hospitalizations (0, 1, 2 or more) | | | | | | |
| < 1; n (%) | 42,437 (67.2%) | 10,868 (74.3%) | -7.1% (-7.9%, -6.3%) | 9,065 (73.5%) | 9,101 (73.8%) | -0.3% (-1.4%, 0.8%) |
| 1 - <2; n (%) | 11,810 (18.7%) | 2,468 (16.9%) | 1.8% (1.1%, 2.5%) | 2,099 (17.0%) | 2,094 (17.0%) | 0.0% (-0.9%, 1.0%) |
| >= 2; n (%) | 8,944 (14.2%) | 1,299 (8.9%) | 5.3% (4.7%, 5.8%) | 1,175 (9.5%) | 1,144 (9.3%) | 0.3% (-0.5%, 1.0%) |
| Heart failure hospitalization; n (%) | 8,052 (12.7%) | 1,429 (9.8%) | 3.0% (2.4%, 3.5%) | 1,191 (9.7%) | 1,216 (9.9%) | -0.2% (-1.0%, 0.5%) |
| ED visit; n (%) | 31,534 (49.9%) | 6,284 (42.9%) | 7.0% (6.1%, 7.9%) | 5,393 (43.7%) | 5,341 (43.3%) | 0.4% (-0.8%, 1.7%) |
| Acute MI; n (%) | 1,567 (2.5%) | 346 (2.4%) | 0.1% (-0.2%, 0.4%) | 297 (2.4%) | 279 (2.3%) | 0.1% (-0.2%, 0.5%) |
| Old MI; n (%) | 5,115 (8.1%) | 1,206 (8.2%) | -0.1% (-0.6%, 0.4%) | 957 (7.8%) | 997 (8.1%) | -0.3% (-1.0%, 0.4%) |
| Heart failure; n (%) | 14,709 (23.3%) | 3,175 (21.7%) | 1.6% (0.8%, 2.3%) | 2,573 (20.9%) | 2,613 (21.2%) | -0.3% (-1.3%, 0.7%) |
| Acute heart failure; n (%) | 5,350 (8.5%) | 982 (6.7%) | 1.8% (1.3%, 2.2%) | 815 (6.6%) | 815 (6.6%) | 0.0% (-0.6%, 0.6%) |
| Microalbuminuria or proteinuria; n (%) | 2,378 (3.8%) | 685 (4.7%) | -0.9% (-1.3%, -0.5%) | 544 (4.4%) | 543 (4.4%) | 0.0% (-0.5%, 0.5%) |
| Dual status/Low income subsidy; n (%) | 20,191 (32.0%) | 3,108 (21.2%) | 10.7% (10.0%, 11.5%) | 2,876 (23.3%) | 2,843 (23.0%) | 0.3% (-0.8%, 1.3%) |
| Ratio of brand to generic medications | | ļ | | | | |
| mean (sd) | 1.02 (0.04) | 1.02 (0.04) | -0.00 (-0.00, -0.00) | 1.02 (0.04) | 1.02 (0.04) | 0.00 (-0.00, 0.00) |
| median [IQR] | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.04] | - (-, -) | 1.00 [1.00, 1.04] | 1.00 [1.00, 1.04] | - (-, -) |
| min, max | 0.83, 1.50 | 0.86, 1.48 | - (-, -) | 0.89, 1.43 | 0.86, 1.48 | - (-, -) |

Variable\_name Algorithm sources Age Gender Race If region not available, from State, https://www2.census.gov/geo/pdfs/mapsdata/maps/reference/us\_regdiv.pdf Region https://www.cms.gov/medicare-medicaid-coordination/medicare-and-medicaidcoordination/medicare-medicaid-coordination-Dual status/Low income subsidy office/downloads/mmco\_dualeligibledefinition.pdf Investigator review of codes based on:  $\underline{https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-projects/AP/repos/sentinel-anal$ packages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002, https://pubmed.ncbi.nlm.nih.gov/34953068/, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9154288/, Smoking / Tobacco use https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3721171/ Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ Underweight Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ Normal weight, if BMI is 20.0-24.9 Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ Overweight, if BMI is 25.0 to 29.9 Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ Class 1 (low-risk) obesity, if BMI is 30.0 to 34.9 Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ Class 2 (moderate-risk) obesity, if BMI is 35.0 to 39.9 Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ Class 3 (high-risk) obesity if BMI is equal to or greater than 40 Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ Unspecified obesity Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/, Diabetic retinopathy https://pubmed.ncbi.nlm.nih.gov/35043165/ Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/, Diabetic neuropathy https://pubmed.ncbi.nlm.nih.gov/35043165/ Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/ Diabetic nephropathy Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/, Diabetes with other opthalmic complications ICD9 to ICD10 conversion Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/books/NBK368403/table/sb203.t5/, https://www.health.mil/Reference-Center/Publications/2016/03/01/Diabetes-Mellitus, http://www.icd9data.com/2014/Volume1/240-279/249-259/250/default.htm, https://www.icd10data.com/ICD10CM/Codes/E00-E89/E08-E13/E11-Diabetes with peripheral circulatory disorders Investigator review of codes based on: (modified codes) Diabetic foot https://pubmed.ncbi.nlm.nih.gov/36102675/ Investigator review of codes based on: the paper then used ICD9/ICD10 website to expand it, https://www.icd10data.com/ICD10CM/Codes/N00-N99/N40-N53/N52-, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4857901/ Erectile dysfuntion Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/, Hypoglycemia https://pubmed.ncbi.nlm.nih.gov/35043165/ Investigator review of codes based on: Hyperglycemia: https://pubmed.ncbi.nlm.nih.gov/34953068/, https://pubmed.ncbi.nlm.nih.gov/35043165/ DKA: https://pubmed.ncbi.nlm.nih.gov/29773640/, https://pubmed.ncbi.nlm.nih.gov/38262528/ HONK:  $\underline{https://dam.assets.ohio.gov/image/upload/medicaid.ohio.gov/Providers/PaymentInnova}$ Hyperglycemia/DKA/HONK tion/DFF/DKA ndf Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/,

ICD9 to ICD10 conversion

Skin infections

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/19337843/, https://pmc.ncbi.nlm.nih.gov/articles/PMC9172873/ Stable angina Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/19337843/, Unstable angina https://pmc.ncbi.nlm.nih.gov/articles/PMC9172873/ Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8929186/ Hypertension Investigator review of codes based on: Hypotension https://pmc.ncbi.nlm.nih.gov/articles/PMC8064679/ Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-Hyperlipidemia packages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015 Atrial fibrillation Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/31933524/ Acute myocardial infarction Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/24682186/ Old myocardial infarction Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/24682186/ Investigator review of codes based on: https://stacks.cdc.gov/view/cdc/31381/cdc\_31381\_DS8.pdf, https://www.health.ny.gov/health\_care/medicaid/redesign/dsrip/vbp\_library/docs/arrblk. pdf, https://www.cdc.gov/dhdsp/maps/atlas/data-sources.html, https://www.cms.gov/medicare/coding/icd10/downloads/icd10clinicalconcepts cardiology1.pdf, ICD9 to ICD10 conversion Cardiac conduction disorder Modified codes based on eligibility criteria, here we implement any care setting, any Previous cardiac procedure (CABG, PTCA, Stent) diagnosis position Modified codes based on eligibility criteria, here we implement any care setting, any Ischemic stroke diagnosis position Investigator review of codes, https://www.icd10data.com/ PVD diagnosis or surgery Investigator review of codes based on: https://stacks.cdc.gov/view/cdc/31381/cdc\_31381\_DS8.pdf, https://www.health.ny.gov/health\_care/medicaid/redesign/dsrip/vbp\_library/docs/arrblk. pdf, https://www.cdc.gov/dhdsp/maps/atlas/data-sources.html, https://www.cms.gov/medicare/coding/icd10/downloads/icd10clinicalconcepts cardiology1.pdf, ICD9 to ICD10 conversion Other cardiac dysrhythmia Modified codes based on inclusion criteria, here we implement any care setting, any Heart failure diagnosis position Modified codes based on inclusion criteria, here we implement any care setting, any Acute heart failure diagnosis position Modified codes based on inclusion criteria, here we implement any care setting, any Microalbuminuria/proteinuria diagnosis position Investigator review of codes based on: https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-Cardiomyopathy packages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015 Investigator review of codes based on: https://stacks.cdc.gov/view/cdc/31381/cdc\_31381\_DS8.pdf, https://pubmed.ncbi.nlm.nih.gov/38440888/, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8751938/, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-Valve disorders packages/browse?at=cder\_mpl2p\_wp009 Modified codes based on eligibility criteria, here we implement any care setting, any Valve replacement diagnosis position Modified codes based on eligibility criteria, here we implement any care setting, any TIA diagnosis position Investigator review of codes based on: https://www.cms.gov/medicare-coveragedatabase/view/article.aspx?articleid=52993&ver=45& Edema Investigator review of codes based on:

https://www.sciencedirect.com/science/article/pii/S2666572723000251

Venous thromboembolism/ pulmonary embolsim

Pulmonary hypertension Investigator review of codes Modified codes based on eligibility criteria, here we implement any care setting, any Implantable cardioverter defibrillator diagnosis position https://pmc.ncbi.nlm.nih.gov/articles/PMC4399109/ Hyperkalemia Investigator review of codes based on: Coronary atherosclerosis https://pmc.ncbi.nlm.nih.gov/articles/PMC10251803/ Cerebrovascular procedure Investigator review of codes, https://www.icd10data.com/ Modified codes based on eligibility criteria, here we implement any care setting, any Insertion of pacemakers / removal of cardiac lead diagnosis position CKD stage 1-2 Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/ Investigator review of codes based on: https://pmc.ncbi.nlm.nih.gov/articles/PMC2978782/ CKD stage 3-4 Investigator review of codes based on: Unspecified CKD https://pmc.ncbi.nlm.nih.gov/articles/PMC5888226/ Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8929186/ Acute kidney injury Investigator review of codes based on: https://nccd.cdc.gov/ckd/Methods.aspx?Qnum=Q637, https://www.kidneymedicinejournal.org/cms/10.1016/j.xkme.2022.100414/attachment/ 5e29ab67-7a7d-4621-9af3-81bd071bbc67/mmc1.pdf, https://www.icd10data.com/ICD10CM/Codes/I00-I99 Hypertensive nephropathy Investigator reviewed code based on: Urinary tract infections  $\underline{https://pmc.ncbi.nlm.nih.gov/articles/PMC7558992/\#app1-antibiotics-09-00536}$ Genital infections Investigator reviewed codes based on: https://pubmed.ncbi.nlm.nih.gov/30207042/ Investigator review of codes based on: Urolithiasis (kidney or urinary stones) https://pmc.ncbi.nlm.nih.gov/articles/PMC7793999/ Investigator review of codes based on: COPD https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10203971/ Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10203971/, modified CCW algorithm Asthma (any care setting, any diagnosis position) Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8636332/, Obstructive sleep apnea https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7927325/ https://pubmed.ncbi.nlm.nih.gov/29921683/, https://pubmed.ncbi.nlm.nih.gov/17346615/, Serious bacterial infections https://pubmed.ncbi.nlm.nih.gov/23335588/ Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10203971/ Pneumonia https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015, Modified algorightm from Liver disease https://pubmed.ncbi.nlm.nih.gov/34256144/, Modified CCW algorithm Investigator review of codes: https://pubmed.ncbi.nlm.nih.gov/32300995/, MASH/MASLD https://pubmed.ncbi.nlm.nih.gov/39316292/ https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=cder\_mpl2p\_wp009, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-Fractures / Falls packages/browse?at=cder\_mpl2p\_wp010 https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8202643/, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic $packages/browse? at \verb|=refs| \% 2 Fheads| \% 2 Fcder\_sir\_wp002, CCW Algorithms|$ Osteoporosis Osteoarthritis Modified CCW algorithm

https://pubmed.ncbi.nlm.nih.gov/35043165/, CCW Algorithms

Depression

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-Dementia

packages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015 https://pubmed.ncbi.nlm.nih.gov/28485014/,

https://pubmed.ncbi.nlm.nih.gov/35043165/,

https://pubmed.ncbi.nlm.nih.gov/35043165/ https://pubmed.ncbi.nlm.nih.gov/35043165/

Investigator review of codes based on https://www.verywellhealth.com/sleeping-disorders-list-

and-diagnostic-codes-3014779

Modified codes based on eligibility criteria, here we implement any care setting, any

diagnosis position

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/38556924/

https://pubmed.ncbi.nlm.nih.gov/34913208/,

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8427377/

Investigator review of codes based on: https://www.cms.gov/icd10m/version37-fullcode-

cms/fullcode\_cms/P0244.html Investigator review of codes based on:

https://pmc.ncbi.nlm.nih.gov/articles/PMC10478599/

Investigator review of codes based on: https://nccd.cdc.gov/ckd/Methods.aspx?Onum=0637.

https://www.cms.gov/icd10m/FY2024-nprmversion41.0-fullcode-

cms/fullcode\_cms/P2401.html

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/38527324/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/37796527/,

https://pubmed.ncbi.nlm.nih.gov/35851329/,

https://pmc.ncbi.nlm.nih.gov/articles/PMC3985913/,

https://pubmed.ncbi.nlm.nih.gov/38503905/, https://pubmed.ncbi.nlm.nih.gov/35513234/

Investigator review of codes: https://pubmed.ncbi.nlm.nih.gov/36222554/,

https://pubmed.ncbi.nlm.nih.gov/30287807/, https://pubmed.ncbi.nlm.nih.gov/22262606/

Investigator review of codes based on: <a href="https://pubmed.ncbi.nlm.nih.gov/36798959/">https://pubmed.ncbi.nlm.nih.gov/36798959/</a>,

https://pubmed.ncbi.nlm.nih.gov/28438588/, https://pubmed.ncbi.nlm.nih.gov/31095068/

Investigator review of codes: https://pubmed.ncbi.nlm.nih.gov/34624355/

Investigator review of codes

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK518983/ Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK278938/

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK513225/ Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK542331/

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK576405/ Investigator review of codes, https://www.drugs.com,

https://www.ncbi.nlm.nih.gov/books/NBK551656/, https://pmc.ncbi.nlm.nih.gov/articles/PMC4882495/,

https://www.ncbi.nlm.nih.gov/books/NBK557848/

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK518983/

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK278938/ Investigator review of codes, https://www.drugs.com,

https://www.ncbi.nlm.nih.gov/books/NBK513225/ Investigator review of codes, https://www.drugs.com,

https://www.ncbi.nlm.nih.gov/books/NBK542331/ Investigator review of codes, https://www.drugs.com,

https://www.ncbi.nlm.nih.gov/books/NBK576405/

Delirium or psychosis

Anxiety

Sleep disorder

Anemia

Influenza

COVID-19

Hyperthyroidism and other thyroid gland disorders

Hypothyroidism

Nephrotic syndrome Urinary incontinence

Biliary disease

Pancreatitis

Bowel obstruction Gastroparesis

Number of antidiabetic drugs on CED

Concomitant use or initiation of metformin

Concomitant use or initiation of insulin

Concomitant use or initiation of sulfonylureas

Concomitant use or initiation of DPP4i

Concomitant use or initiation of SGLT2i

Concomitant use or initiation of other glucose-lowering drugs

Past use of metformin

Past use of insulin

Past use of sulfonylureas

Past use of DPP4i

Past use of SGLT2i

https://www.ncbi.nlm.nih.gov/books/NBK551656/, https://pmc.ncbi.nlm.nih.gov/articles/PMC4882495/, Past use of other glucose-lowering drugs https://www.ncbi.nlm.nih.gov/books/NBK557848/ Investigator review of codes, https://www.drugs.com, ACEi / ARB https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/ Investigator review of codes, https://www.drugs.com, ARNI https://www.ncbi.nlm.nih.gov/books/NBK507904/ Investigator review of codes, https://www.drugs.com, Thiazides https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/ Investigator review of codes, https://www.drugs.com, Beta-Blockers https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/ Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/ Calcium channel blockers Investigator review of codes, https://www.drugs.com. https://www.ncbi.nlm.nih.gov/books/NBK556025/, Digoxin / Digitoxin https://pubchem.ncbi.nlm.nih.gov/compound/441207 Investigator review of codes, https://www.drugs.com, Loop diuretics https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/ Investigator review of codes, https://www.drugs.com, Other diuretics https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/ Intravenous diuretics Investigator review of codes Investigator review of codes, https://www.drugs.com, Nitrates https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/ Investigator review of codes, https://www.drugs.com,  $https://www.ncbi.nlm.nih.gov/books/NBK482322/ \, (using \, class \, I \, and \, class \, II \, as \, class \, 2 \, is \, (using \, class \, I) \, (using \, class \, I)$ Anti-arrhythmics beta blockers and class 4 is calcium channel blockers) Investigator review of codes, https://www.drugs.com, https://www.heart.org/en/health- $\underline{topics/cholesterol/prevention-and-treatment-of-high-cholesterol-}$ Statins hyperlipidemia/cholesterol-medications Investigator review of codes, https://www.drugs.com, https://www.heart.org/en/healthtopics/cholesterol/prevention-and-treatment-of-high-cholesterol-PCSK9 inhibitors and other lipid-lowering drugs <u>hyperlipidemia/cholesterol-medications</u> Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK537062/ Antiplatelet agents Investigator review of codes, https://www.drugs.com, Oral anticoagulants https://www.ahajournals.org/doi/full/10.1161/JAHA.120.017559 Investigator review of codes, https://www.copdfoundation.org/Learn-More/I-am-a-Person-with-COPD/Treatments-Medications.aspx, COPD/Asthma medication https://getasthmahelp.org/medications-list.aspx Investigator review of codes, https://www.drugs.com, **NSAIDs** https://www.ncbi.nlm.nih.gov/books/NBK547742/ Investigator review of codes, https://www.drugs.com, https://www.aaaai.org/tools-for-Oral corticosteroids the-public/drug-guide/oral-corticosteroid-medications Investigator review of codes based on: https://www.drugs.com. Osteoporosis agents (incl. bisphosphonates) https://www.ncbi.nlm.nih.gov/books/NBK470248/ Investigator review of codes, https://www.drugs.com, https://pubmed.ncbi.nlm.nih.gov/31643200/#:~:text=They%20can%20also%20be%20i Opioids nformally,%2C%20codeine%2C%20oxycodone%2C%20hydrocodone%2C Investigator review of codes, https://www.drugs.com, Anti-depressants https://www.ncbi.nlm.nih.gov/books/NBK538182/ Antipsychotics Investigator review of codes, https://www.drugs.com Investigator review of codes, https://www.drugs.com, https://www.dea.gov/sites/default/files/2020-06/Benzodiazepenes-2020.pdf, Anxiolytics/hypnotics, benzodiazepines https://www.ncbi.nlm.nih.gov/books/NBK470159/, https://www.drugs.com Investigator review of codes based on: https://www.drugs.com,

Medication for dementia

Urinary tract infections antibiotics

Number of distinct medications, median (iqr), mean (sd)

Investigator review of codes, https://www.drugs.com,

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7462122/,

https://go.drugbank.com/drugs/DB00382

https://pubmed.ncbi.nlm.nih.gov/35790044/ Investigator review of codes, https://www.drugs.com

https://www.cms.gov/files/document/mm13473-how-use-office-and-outpatientevaluation-and-management-visit-complexity-add-code-g2211.pdf, https://www.cms.gov/files/document/physician-fee-schedule-pfs-paymentofficeoutpatient-evaluation-and-management-em-visits-fact-sheet.pdf Number of office visits median (igr), mean (sd) Data dictionary of Optum, Marketscan and https://www.cms.gov/Medicare/Provider-Enroll ment- and - Certification / Medicare Provider Sup Enroll / downloads / taxonomy.pdf,https://www.cms.gov/medicare/provider-enrollment-and-Number of endocrinologist visits, median (iqr), mean (sd) certification/medicareprovidersupenroll/downloads/taxonomycrosswalk.pdf Data dictionary of Optum, Marketscan and https://www.cms.gov/Medicare/Provider-Enrollment-and-Certification/MedicareProviderSupEnroll/downloads/taxonomy.pdf. https://www.cms.gov/medicare/provider-enrollment-andcertification/medicareprovidersupenroll/downloads/taxonomycrosswalk.pdf Number of cardiologist visits, median (iqr), mean (sd) Data dictionary of Optum, Marketscan and https://www.cms.gov/Medicare/Provider-Enrollment-and-Certification/MedicareProviderSupEnroll/downloads/taxonomy.pdf, https://www.cms.gov/medicare/provider-enrollment-andcertification/medicareprovidersupenroll/downloads/taxonomycrosswalk.pdf Number of internal medicine/family medicine visits, median (iqr), mean (sd) https://www.cms.gov/medicare-coverage-database/view/article.aspx?articleId=57326, https://firstcoastbillinggroup.com/ekg-billing-and-reimbursement/, https://www.aapc.com/codes/coding-newsletters/my-cardiology-coding-alert/cpt-Number of electrocardiograms, median (iqr), mean (sd) answer-5-common-ecg-coding-questions-175952-article https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8511132/,https://pubmed.ncbi.nlm.nih.gov/34778785/, https://www.cms.gov/medicare-coveragedatabase/view/article.aspx?articleid=56625&ver=27&, https://www.medicalbillgurus.com/echocardiogram-cpt-code/ Number of echocardiograms, median (iqr), mean (sd) Pharmacy out-of-pocket cost, median (igr), mean (sd) Investigator review of codes, https://www.drugs.com Unique brand medications Investigator review of codes, https://www.drugs.com Unique generic medications Ratio of unique brand to generic medications Investigator review of codes, https://www.drugs.com https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-Colonoscopy/ Sigmoidoscopy packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002 nttps://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002, https://www.cms.gov/medicare-coveragedatabase/view/article.aspx?articleId=54767&DocID=A54767, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002, https://www.cms.gov/medicare-coveragedatabase/view/article.aspx?articleId=54767&DocID=A54767 Flu vaccine / Pneumococcal vaccine https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002, http://www.icd9data.com/2012/Volume1/V01-V91/V70-V82/V72/default.htm, Pan smear test http://www.icd9data.com/2012/Volume1/V01-V91/V70-V82/V76/default.htm https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-PSA test packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002 Fecal occult blood test Investigator review of codes Bone mineral density tests Investigator review of codes based on: https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002. https://www.cms.gov/medicare-coveragedatabase/view/article.aspx?articleid=56448&ver=16&bc=0, http://www.icd9data.com/2012/Volume1/V01-V91/V70-V82/V76/default.htmMammograms Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/33151319/, https://www.cms.gov/newsroom/fact-sheets/medicare-telemedicine-health-care-provider-fact-sheets/medicare-provider-fact-sheets/medicare-fact-sheets/medicar sheet, https://www.aafp.org/family-physician/practice-and-career/getting-paid/coding/coding-Telemedicine telehealth-audio-virtual-digital-visits.html Number of HbA1c tests, median (iqr), mean (sd) https://pubmed.ncbi.nlm.nih.gov/34953068/ Number of lipid panels, median (igr), mean (sd) https://pubmed.ncbi.nlm.nih.gov/34953068/ https://pubmed.ncbi.nlm.nih.gov/34953068/ Number of creatinine tests, median (igr), mean (sd)

Investigator review of codes

Investigator review of codes

N/A

Number of natriuretic peptide tests, median (iqr), mean (sd)

Number of urine tests, median (iqr), mean (sd)

HbA1c

Glucose N/A Creatinine N/A Systolic blood pressure N/A Heart rate N/A ВМІ N/A eGFR N/A LDL N/A HDL N/A Total cholesterol N/A Triglycerides N/A

Combined comorbidity score

Frailty score

Number of any hospitalization, median (iqr), mean (sd)

Any hospitalization within prior 90 days; n (%)

Any hospitalization within prior 91-365 days; n (%)

N/A

0,1, >1 hospitalizations (any)

Hospitalization for heart failure; n (%)

N/A

Different in all 3 databases and measure already created in all 3 as well;

 $ED\ visit\ (Medicare): Revenue\ center\ codes:\ 0450,0451,0452,0456,0459,0981; Place$ 

 $\underline{\textbf{A combined comorbidity score predicted mortality in elderly patients better than}$ 

Measuring Frailty in Medicare Data: Development and Validation of a Claims-Based

existing scores, https://pubmed.ncbi.nlm.nih.gov/21208778/

Frailty Index, https://pubmed.ncbi.nlm.nih.gov/29244057/

of service: 23

ED visit (Optum): Place of service: 23

ED visit (Marketscan): Service sub-category codes: 10120, 10220, 10320, 10420, 10520, 12220, 20120, 20220, 21120, 21220, 22120, 22320, 30120, 30220, 30320, 30420, 30520, 30620, 31120, 31220, 31320, 31420, 31520, 31620; Place of service: 23

20, 30020, 31120, 31220, 3132

Number of emergency department visit median (iqr), mean (sd)

Calendar year

N/A

## TIRZSEMA-CVOT-TIRZDULA

## **Appendices**

- 1 Target Trial Framework, Operational Definitions and Data Fitness Assessment
- 2 Code algorithms
- 2a Exposure
- 2b Inclusion
- 2c Exclusion
- 2d Outcome
- 3 Flowchart for cohort assembly
- 4 1st feasibility assessment
- 5 2nd feasibility assessment
- 6 Balance Assessment PS Distribution and C-Statistic
- 7 Balance Assessment Table 1
- 8 Covariate Algorithm Sources

| | TIRZDULA | OPTUM | MARKETSCAN | Notes/Questions | Color coding |
|---|---|---|---|---|---|
| | International, double-blind, randomized, active- | Non-randomized initiation of treatment Tirzepatide vs Dulaglutide | Non-randomized initiation of treatment Tirzepatide vs Dulaglutide | | |
| index date) | controlled trial to treatment A vs B | (first eligible entry to study population) | (first eligible entry to study population) | | Good proxy definition |
| | | Code type: RX Care setting: N/A | Code type: RX Care setting: N/A | | |
| | | Diagnosis position: N/A | Diagnosis position: N/A | | |
| | | Washout window: [-183,-1] Incident with respect to: Tirzepatide in any formulation or dose | Washout window: [-183, -1] Incident with respect to: Tirzepatide in any formulation or dose | | |
| | | Assessment window: N/A | Assessment window: N/A | | |
| | Tirzepatide (subcutaneously once per week) | Source of algorithm: N/A Measurement characteristics: N/A | Source of algorithm: N/A Measurement characteristics: N/A | | Moderate proxy definition |
| Exposure | once per week) | Code type: RX | Code type: RX | | Moderate proxy definition |
| | | Care setting: N/A Diagnosis position: N/A | Care setting: N/A Diagnosis position: N/A | | |
| | | Washout window: [-183, -1] | Washout window: [-183, -1] | | |
| | | Incident with respect to: Dulaglutide in any formulation or dose | Incident with respect to: Dulaglutide in any formulation or dose | | |
| | | Assessment window: N/A Source of algorithm: N/A | Assessment window: N/A Source of algorithm: N/A | | |
| Comparator | Dulaglutide (subcutaneously once per week) | Measurement characteristics: N/A | Measurement characteristics: N/A | | Poorly measured in database |
| | | Code type: DX, PX Care setting: Inpatient for stroke/MI, any for death | Code type: DX, PX Care setting: Inpatient for stroke/MI, any for death | | |
| | | Diagnosis position: Primary for Stroke, Any for MI | Diagnosis position: Primary | | |
| | | Washout window: Source of algorithm: Measurement characteristics: Death includes information | Washout window: Source of algorithm: Measurement characteristics: Death includes information | | |
| | | from the inpatient discharged dead status, social security death master file, and | from the inpatient discharged dead status, social security death master file, and | | Poorly measured in database and no |
| Primary outcome to be emulated | MACE, defined as CV death, MI, or stroke | deaths scraped from obituaries or other sources. Code type: DX. PX | deaths scraped from obituaries or other sources. Code type: DX, PX | | important |
| | | Care setting: Inpatient for stroke/MI/ heart failure, any for death, outpatient for i.v. | Care setting: Inpatient for stroke/MI/ heart failure, any for death, outpatient for i.v. | | |
| | | diuretics Diagnosis position: Primary for stroke/ heart failure, any for MI | diuretics Diagnosis position: Primary for stroke/ heart failure, any for MI | | |
| | | Washout window: | Washout window: | | |
| | | Source of algorithm: PROMISE Team, Validation studies, (Investigator reviewed codes) | Source of algorithm: PROMISE Team, Validation studies, (Investigator reviewed codes) | | |
| | | Measurement characteristics: Death includes information from the inpatient | Measurement characteristics: Death includes information from the inpatient | | |
| | | discharged dead status, social security death master file, and deaths scraped from obituaries or other sources. | discharged dead status, social security death master file, and deaths scraped from obituaries or other sources. | | |
| | | PPV for ischemic stroke using ICD9 codes was 88% and 95% | PPV for ischemic stroke using ICD9 codes was 88% and 95% | | |
| | | [https://pubmed.ncbi.nlm.nih.gov/12364739/ and<br>https://pubmed.ncbi.nlm.nih.gov/20140892/] | [https://pubmed.ncbi.nlm.nih.gov/12364739/ and<br>https://pubmed.ncbi.nlm.nih.gov/20140892/] | | |
| | | Both of the above ICD9 codes were mapped to ICD10, but no validation study was | Both of the above ICD9 codes were mapped to ICD10, but no validation study was | | |
| | all-cause mortality, myocardial infarction, or stroke. | performed. PPV for HHF diagnosis using ICD-10 codes was 98% in a national Medicare. | performed. PPV for HHE diagnosis using ICD-10 codes was 98% in a national Medicare. | | |
| | heart failure, or urgent heart failure visits requiring | sample. | sample. | | |
| emulated | intravenous diuretics.<br>Randomization date | One day after initiation of treatment with tirzepatide or dulaglutide | One day after initiation of treatment with tirzepatide or dulaglutide | | |
| rollow up start | Nandomization date | Earliest of: Outcome, end of observation in data, end of study period (365 days), | Earliest of: Outcome, end of observation in data, end of study period (365 days), | | |
| Follow up end | 1. com | discontinuation of study drug (45 days grace window and risk-window), switch to other GLP-1-RA, nursing home admission | discontinuation of study drug (45 days grace window and risk-window), switch to other GLP-1-RA, nursing home admission | | |
| rollow up end | 1 year | other GEP-1-NA, hursing home authission | other GEF-1-RA, hursing nome aurilission | Algorithm detail: Adherence in clinical practice databases is | |
| | | | | expected to be much worse than in the trial, therefore the on-<br>treatment analysis at 1 year follow-up will be the primary | |
| Causal estimand | Intention-to-treat effect | On-treatment effect | On-treatment effect | analysis. | |
| Effect estimation<br>Inclusion criteria | Cox proportional hazards model | Cox proportional hazards regression model | Cox proportional hazards regression model | | |
| inclusion criteria | | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | | |
| | | Assessment window: [0, 0] Code type: N/A | Assessment window: [0, 0] Code type: N/A | | |
| | | Care setting: N/A | Caresetting: N/A | | |
| | | Diagnosis position: N/A | Diagnosis position: N/A | | |
| 1 | Men and women aged 18 years or older | Source of algorithm: N/A Measurement characteristics: N/A | Source of algorithm: N/A Measurement characteristics: N/A | | |
| | | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | | |
| | | Assessment window: [-365, 0] Code type: DX | Assessment window: [-365, 0] Code type: DX | | |
| | | Care setting: Any | Care setting: Any | | |
| | | Diagnosis position: Any Source of algorithm: PROMISE team | Diagnosis position: Any Source of algorithm: PROMISE team | | |
| 2 | Type 2 diabetes mellitus | Measurement characteristics: N/A | Measurement characteristics: N/A | | |
| | | Applied before/after selection of index date: Before Assessment window: [-730, 0] | Applied before/after selection of index date: Before Assessment window: [-730, 0] | | |
| | | Code type: DX, LOINC | Code type: DX, LOINC | | |
| | | Care setting: Any Diagnosis position: Any | Care setting: Any Diagnosis position: Any | | |
| | | Source of algorithm: Validation of obesity-related diagnosis codes in claims | Source of algorithm: Validation of obesity-related diagnosis codes in claims | | |
| | | data: Validation of body mass index (BMI)-related ICD-9-CM and ICD-10-CM administrative diagnosis codes recorded in US claims data | data; Validation of body mass index (BMI)-related ICD-9-CM and ICD-10-CM administrative diagnosis codes recorded in US claims data | Algorithm detail: If BMI measurement via LOINC code is | |
| | $BMI \ge 25kg/m2$ | Measurement characteristics: N/A | Measurement characteristics: N/A | below 10 or above 100 then measurent is set to missing. | |
| | Low, moderate, or high cardiovascular risk, definde<br>History of a cardiovascular event | ed as either one of: | | | |
| 4.1 | or a cardiovascuidi everit | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | | |
| | | Assessment window: [all available data, 0] Code type: DX | Assessment window: [all available data, 0] Code type: DX | | |
| | | Care setting: Any | Care setting: Any | | |
| | Decrimented history of my condictinfore* | Diagnosis position: Any Source of algorithm: N/A | Diagnosis position: Any Source of algorithm: N/A | | |
| 4.1.1 | Documented history of myocardial infarction or<br>unstable angina | Source of algorithm: N/A Measurement characteristics: N/A | Source of algorithm: N/A Measurement characteristics: N/A | | |

easured in database and not

| | | Applied before/after selection of index date: Before Assessment window: [all available data, 0] | Applied before/after selection of index date: Before Assessment window: [all available data, 0] |
|---|---|---|---|
| | | Code type: DX | Code type: DX |
| | | Care setting: Any | Care setting: Any |
| | | Diagnosis position: Any | Diagnosis position: Any |
| | | Source of algorithm: N/A | Source of algorithm: N/A |
| 4.1.2 | History of ischemic stroke or TIA | Measurement characteristics: N/A Applied before/after selection of index date: Before | Measurement characteristics: N/A Applied before/after selection of index date: Before |
| | | Assessment window: [all available data, 0] | Assessment window: [all available data, 0] |
| | | Code type: DX | Code type: DX |
| | | Care setting: Any | Care setting: Any |
| | | Diagnosis position: Any | Diagnosis position: Any |
| | | Source of algorithm: DUPLICATE team, investigator reviewed codes | Source of algorithm: DUPLICATE team, investigator reviewed codes |
| 4.1.3 | History of heart failure | Measurement characteristics: N/A | Measurement characteristics: N/A |
| | | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before |
| | | Assessment window: [all available data, 0] Code type: DX | Assessment window: [all available data, 0] Code type: DX |
| | | Care setting: Any | Care setting: Any |
| | | Diagnosis position: Any | Diagnosis position: Any |
| | History of surgical or percutaneous coronary | Source of algorithm: PROMISE team | Source of algorithm: PROMISE team |
| 4.1.4 | revascularization procedure | Measurement characteristics: N/A | Measurement characteristics: N/A |
| | | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before |
| | | Assessment window: [all available data, 0] Code type: DX, PX | Assessment window: [all available data, 0] Code type: DX, PX |
| | | Care setting: Any | Caresetting: Any |
| | | Diagnosis position: Any | Diagnosis position: Any |
| | History of carotid stenting or surgical | Source of algorithm: N/A | Source of algorithm: N/A |
| 4.1.5 | revascularization | Measurement characteristics: N/A | Measurement characteristics: N/A |
| | | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before |
| | | Assessment window: [all available data, 0] | Assessment window: [all available data, 0] |
| | | Code type: DX, PX | Code type: DX, PX<br>Care setting: Any |
| | | Care setting: Any Diagnosis position: Any | Diagnosis position: Any |
| | History of peripheral vascular procedure (stenting or | Source of algorithm: N/A | Source of algorithm: N/A |
| 4.1.6 | surgical revascularization) | Measurement characteristics: N/A | Measurement characteristics: N/A |
| | , | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before |
| | | Assessment window: [all available data, 0] | Assessment window: [all available data, 0] |
| | | Code type: RX | Code type: RX |
| | | Care setting: N/A Diagnosis position: N/A | Care setting: N/A Diagnosis position: N/A |
| | | Source of algorithm: Primary agents as defined by ACC/AHA guidelines for high. | Source of algorithm: Primary agents as defined by ACC/AHA guidelines for high |
| | | blood pressure | blood pressure |
| 4.2 | Current use of ≥1 antihypertensive drug | Measurement characteristics: N/A | Measurement characteristics: N/A |
| | | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before |
| | | Assessment window: [all available data, 0] | Assessment window: [all available data, 0] |
| | | Code type: RX | Code type: RX |
| | | Care setting: N/A Diagnosis position: N/A | Care setting: N/A Diagnosis position: N/A |
| | | Source of algorithm: Common lipid-lowering medications as defined by | Source of algorithm: Common lipid-lowering medications as defined by |
| | | ACC/AHA guidelines on management of blood cholesterol | ACC/AHA guidelines on management of blood cholesterol |
| 4.3 | Current use of ≥1 lipid-lowering drug | Measurement characteristics: N/A | Measurement characteristics: N/A |
| | | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before |
| | | Assessment window: [all available data, 0] | Assessment window: [all available data, 0] |
| | | Code type: DX | Code type: DX |
| | | Care setting: Any Diagnosis position: Any | Caresetting: Any Diagnosis position: Any |
| | | Source of algorithm: N/A | Source of algorithm: N/A |
| 4.4.1 | Documented history of coronary artery disease | Measurement characteristics: N/A | Measurement characteristics: N/A |
| | | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before |
| | | Assessment window: [all available data, 0] | Assessment window: [all available data, 0] |
| | | Code type: DX | Code type: DX |
| | | Care setting: Any Diagnosis position: Any | Care setting: Any Diagnosis position: Any |
| | | Source of algorithm: N/A | Source of algorithm: N/A |
| 4.4.2 | Documented history of carotid artery disease | Measurement characteristics: N/A | Measurement characteristics: N/A |
| 7.7.2 | | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before |
| | | Assessment window: [all available data, 0] | Assessment window: [all available data, 0] |
| | | Code type: DX | Code type: DX |
| | | Care setting: Any | Care setting: Any |
| | | Diagnosis position: Any Source of algorithm: N/A | Diagnosis position: Any Source of algorithm: N/A |
| 443 | Documented history of peripheral artery disease | Measurement characteristics: N/A | Measurement characteristics: N/A |
| Exclusion criteria | Decarron and instant of peripheral artery disease | | |
| | | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before |
| | | Assessment window: [-365, 0] | Assessment window: [-365, 0] |
| | | Code type: DX | Code type: DX |
| | | Care setting: Any | Caresetting: Any |
| | | Diagnosis position: Any Source of algorithm: PROMISE team | Diagnosis position: Any Source of algorithm: PROMISE team |
| = | History of T1DM or secondary diabetes | Source of algorithm: PROMISE team Measurement characteristics: N/A | Source of algorithm: PROMISE team Measurement characteristics: N/A |
| 3 | Thistory of 1 10 lvi of secondary diabetes | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before |
| | | Assessment window: [all available data, 0] | Assessment window: [all available data, 0] |
| | | Code type: DX | Code type: DX |
| | | Care setting: Any | Care setting: Any |
| | | Diagnosis position: Any | Diagnosis position: Any |
| ā | Family or personal history of multiple endocrine | Source of algorithm: PROMISE team | Source of algorithm: PROMISE team |
| 6 | neoplasia or medullary thyroid carcinoma | Measurement characteristics: N/A | Measurement characteristics: N/A |

| <b>7</b> End-stage renal disease or dialysis | Applied before/after selection of index date: Before Assessment window: [-365,0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A | Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A | Algorithm detail: Proxied by ICD-10-CM codes for chronic kidney disease stage 5 OR end-stage renal disease OR ICD-10-CM procedure codes for dialysis. |
|---|---|---|---|
| History of treatment for diabetic retinopathy and/or <b>8</b> macular edema | Applied before/after selection of index date: Before Assessment window: [-365,0] Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A | Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A | Algorithm detail: Will be proxied by a history of treatment (e.g. codes for intravitreal injection of anti-VEGFi OR photocoagulation) |
| 9 History of any malignancy | Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: NIA Applied before/after selection of index date: Before Assessment window: [7, 0] | Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [7, 0] | |
| 10 Cardiovascular event or intervention in the past 7 days | Code type: DX, PX Care setting: Inpatient/ED for MI, Stroke, TIA, inpatient for procedures Diagnosis position: Any Source of algorithm: PROMISE team, Investigator reviewed codes Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365,0] Code type: DX Care settins: Any | Code type: DX, PX Care setting: Inpatient/ED for MI, Stroke, TIA, inpatient for procedures Diagnosis position: Any Source of algorithm: PROMISE team, Investigator reviewed codes Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any | |
| 11 Women who are pregnant or breastfeeding | Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [:183, 0] Code type: RX Care setting: N/A Diagnosis position: N/A | Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-183, 0] Code type: RX Care setting: N/A Diagnosis position: N/A | Algorithm detail: Proxied by ICD-10-CM codes indicative of pregnancy at baseline. |
| 12 GLP-1-RA treatment within past 6 months 13 Bariatric surgery within the past 12 months | Source of algorithm: PROMISE team Measurement characteristics: n/a Applied before/after selection of index date: Before Assessment window: [-365, 0] Codet type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A | Source of algorithm:N/A Measurement characteristics: n/a Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A | |


TIA
TIA
TIA
TIA
TIA
TIA
TIA
TIA
TIA


BYPASS CORONARY ARTERY, THREE ARTERIES FROM LEFT


DILATION OF CORONARY ARTERY, TWO ARTERIES, BIFURCATION,


DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION,


DILATION OF CORONARY ARTERY, FOUR OR MORE ARTERIES,


DILATION OF RIGHT COMMON CAROTID ARTERY WITH THREE


DILATION OF LEFT COMMON CAROTID ARTERY WITH THREE


DILATION OF LEFT INTERNAL CAROTID ARTERY WITH THREE


| History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) 0410099 PX WITH AUTOLOGOUS VENOUS TISSUE, OPEN APPROACH | |
|---|---|
| History of peripheral vascular | H ICD-10-PCS |
| procedure (stenting or surgical BYPASS ABDOMINAL AORTA TO LEFT INTERNAL ILIAC 4.1.6 revascularization) 041009B PX AUTOLOGOUS VENOUS TISSUE, OPEN APPROACH History of peripheral vascular | ARTERY WITH ICD-10-PCS |
| procedure (stenting or surgical BYPASS ABDOMINAL AORTA TO BILATERAL INTERNAL 4.1.6 revascularization) 041009C PX ARTERIES WITH AUTOLOGOUS VENOUS TISSUE, OPEN A History of peripheral vascular | |
| procedure (stenting or surgical BYPASS ABDOMINAL AORTA TO RIGHT EXTERNAL ILIA 4.1.6 revascularization) 041009D PX WITH AUTOLOGOUS VENOUS TISSUE, OPEN APPROACH History of peripheral vascular | |
| procedure (stenting or surgical 4.1.6 revascularization) 041009F PX AUTOLOGOUS VENOUS TISSUE, OPEN APPROACH History of peripheral vascular | CARTERY WITH ICD-10-PCS |
| procedure (stenting or surgical BYPASS ABDOMINAL AORTA TO BILATERAL EXTERNA 4.1.6 revascularization) 041009G PX ARTERIES WITH AUTOLOGOUS VENOUS TISSUE, OPEN A History of peripheral vascular | |
| procedure (stenting or surgical BYPASS ABDOMINAL AORTA TO RIGHT FEMORAL ARTE 4.1.6 revascularization) 041009H PX AUTOLOGOUS VENOUS TISSUE, OPEN APPROACH History of peripheral vascular | ERY WITH ICD-10-PCS |
| procedure (stenting or surgical BYPASS ABDOMINAL AORTA TO LEFT FEMORAL ARTEI 4.1.6 revascularization) 041009J PX AUTOLOGOUS VENOUS TISSUE, OPEN APPROACH History of peripheral vascular | RY WITH ICD-10-PCS |
| procedure (stenting or surgical BYPASS ABDOMINAL AORTA TO BILATERAL FEMORAL 4.1.6 revascularization) 041009K PX WITH AUTOLOGOUS VENOUS TISSUE, OPEN APPROACH History of peripheral vascular | |
| procedure (stenting or surgical BYPASS ABDOMINAL AORTA TO LOWER EXTREMITY AI 4.1.6 revascularization) 041009Q PX AUTOLOGOUS VENOUS TISSUE, OPEN APPROACH History of peripheral vascular | RTERY WITH ICD-10-PCS |
| procedure (stenting or surgical BYPASS ABDOMINAL AORTA TO LOWER ARTERY WITH 4.1.6 revascularization) 041009R PX VENOUS TISSUE, OPEN APPROACH History of peripheral vascular | AUTOLOGOUS ICD-10-PCS |
| procedure (stenting or surgical BYPASS ABDOMINAL AORTA TO RIGHT COMMON ILIAC 4.1.6 revascularization) 04100A6 PX AUTOLOGOUS ARTERIAL TISSUE, OPEN APPROACH | ARTERY WITH ICD-10-PCS |
| History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) 04100A7 PX BYPASS ABDOMINAL AORTA TO LEFT COMMON ILIAC A AUTOLOGOUS ARTERIAL TISSUE, OPEN APPROACH | ARTERY WITH ICD-10-PCS |
| History of peripheral vascular procedure (stenting or surgical BYPASS ABDOMINAL AORTA TO BILATERAL COMMON 4.1.6 revascularization) 04100A8 PX ARTERIES WITH AUTOLOGOUS ARTERIAL TISSUE, OPEN | |
| History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) 04100A9 PX WITH AUTOLOGOUS ARTERIAL TISSUE, OPEN APPROACE WITH AUTOLOGOUS ART | |
| History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) 04100AB PX BYPASS ABDOMINAL AORTA TO LEFT INTERNAL ILIAC AUTOLOGOUS ARTERIAL TISSUE, OPEN APPROACH | ARTERY WITH ICD-10-PCS |
| History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) 04100AC PX BYPASS ABDOMINAL AORTA TO BILATERAL INTERNAL ARTERIES WITH AUTOLOGOUS ARTERIAL TISSUE, OPEN | |
| History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) 04100AD PX WITH AUTOLOGOUS ARTERIAL TISSUE, OPEN APPROACH WITH AUTOLOGOUS ART | |
| History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) 04100AF PX BYPASS ABDOMINAL AORTA TO LEFT EXTERNAL ILIAC AUTOLOGOUS ARTERIAL TISSUE, OPEN APPROACH | CARTERY WITH ICD-10-PCS |


| History of peripheral vascular procedure (stenting or surgical DILATION OF LEFT PERONEAL ARTERY, BI 4.1.6 revascularization) 047U066 PX DRUG-ELUTING INTRALUMINAL DEVICES, History of peripheral vascular | |
|---|---|
| procedure (stenting or surgical DILATION OF LEFT PERONEAL ARTERY WI 4.1.6 revascularization) 047U06Z PX INTRALUMINAL DEVICES, OPEN APPROACH History of peripheral vascular | |
| procedure (stenting or surgical DILATION OF LEFT PERONEAL ARTERY, BI 4.1.6 revascularization) 047U076 PX MORE DRUG-ELUTING INTRALUMINAL DEV History of peripheral vascular | |
| procedure (stenting or surgical DILATION OF LEFT PERONEAL ARTERY WI 4.1.6 revascularization) 047U07Z PX ELUTING INTRALUMINAL DEVICES, OPEN A History of peripheral vascular | |
| procedure (stenting or surgical DILATION OF LEFT PERONEAL ARTERY, BI 4.1.6 revascularization) 047U0D6 PX INTRALUMINAL DEVICE, OPEN APPROACH History of peripheral vascular | |
| procedure (stenting or surgical DILATION OF LEFT PERONEAL ARTERY WI 4.1.6 revascularization) 047U0DZ PX OPEN APPROACH History of peripheral vascular | TH INTRALUMINAL DEVICE, ICD-10-PCS |
| procedure (stenting or surgical DILATION OF LEFT PERONEAL ARTERY, BI 4.1.6 revascularization) 047U0E6 PX INTRALUMINAL DEVICES, OPEN APPROACH History of peripheral vascular | |
| procedure (stenting or surgical DILATION OF LEFT PERONEAL ARTERY WI 4.1.6 revascularization) 047U0EZ PX DEVICES, OPEN APPROACH History of peripheral vascular | ITH TWO INTRALUMINAL ICD-10-PCS |
| procedure (stenting or surgical DILATION OF LEFT PERONEAL ARTERY, BI 4.1.6 revascularization) 047U0F6 PX INTRALUMINAL DEVICES, OPEN APPROACH History of peripheral vascular | |
| procedure (stenting or surgical DILATION OF LEFT PERONEAL ARTERY WI 4.1.6 revascularization) 047U0FZ PX DEVICES, OPEN APPROACH | TH THREE INTRALUMINAL ICD-10-PCS |
| History of peripheral vascular procedure (stenting or surgical DILATION OF LEFT PERONEAL ARTERY, BI 4.1.6 revascularization) 047U0G6 PX MORE INTRALUMINAL DEVICES, OPEN API | |
| History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) 047U0GZ PX INTRALUMINAL DEVICES, OPEN APPROAC | |
| History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) 047U0Z6 PX APPROACH | FURCATION, OPEN ICD-10-PCS |
| History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) 047U0ZZ PX DILATION OF LEFT PERONEAL ARTERY, OF | PEN APPROACH ICD-10-PCS |
| History of peripheral vascular procedure (stenting or surgical DILATION OF LEFT PERONEAL ARTERY, BIL 4.1.6 revascularization) 047U346 PX ELUTING INTRALUMINAL DEVICE, PERCUT | , |
| History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) 047U34Z PX INTRALUMINAL DEVICE, PERCUTANEOUS | APPROACH ICD-10-PCS |
| History of peripheral vascular procedure (stenting or surgical DRUG-ELUTING INTRALUMINAL DEVICES, 4.1.6 revascularization) 047U356 PX APPROACH | |
| History of peripheral vascular procedure (stenting or surgical DILATION OF LEFT PERONEAL ARTERY WI 4.1.6 revascularization) 047U35Z PX INTRALUMINAL DEVICES, PERCUTANEOUS | S APPROACH ICD-10-PCS |
| History of peripheral vascular procedure (stenting or surgical 4.1.6 revascularization) HISTORY DELATION OF LEFT PERONEAL ARTERY, BILD DRUG-ELUTING INTRALUMINAL DEVICES, APPROACH | |


| END STAGE RENAL DISEASE (ESRD) RELATED SERVICES DURING THE COURSE OF |
|-----------------------------------------------------------------------------|
| TREATMENT, FOR PATIENTS 20 YEARS OF AGE AND OVER; WITH 1 FACE-TO-FACE |
| PHYSICIAN VISIT PER MONTH / END STAGE RENAL DISEASE (ESRD) RELATED SERVICES |
| DURING THE COURSE OF TREATMENT, FOR PATIENTS 20 YEARS OF AGE AND OVER; WITH |


Compon ent1 overlap with compon ent 2 OR compon ent 3 Compon ent1 overlap with compon ent 2 OR compon ent 3 Compon ent1 overlap with compon ent 2 OR compon ent 3 Compon ent 1 overlap with compon ent 2 OR compon ent 3


| Bariatric s | surgery within the | | GASTRIC RESTRICTIVE PROCEDURE, WITH SMALL INTESTINE RECONSTRUCTION TO | |
|---|---|---|---|---|
| <b>13</b> past 12 m | onths | 43847 PX | LIMIT ABSORPTION; WITH LONG LIMB (>150 CM) ROUX-EN-Y | CPT/HCPCS |
| | surgery within the | | | |
| <b>13</b> past 12 m | onths | 43659 PX | GASTRECTOMY, TOTAL; WITH ROUX-EN-Y RECONSTRUCTION; MINI-GASTRIC BYPASS | CPT/HCPCS |
| Bariatric s | surgery within the | | LAPAROSCOPY, SURGICAL; GASTRIC RESTRICTIVE PROCEDURE, ADJUSTABLE GASTRIC | |
| <b>13</b> past 12 m | onths | S2082 PX | BAND INCLUDES PLACEMENT OF SUBCUTANEOUS PORT | CPT/HCPCS |
| Bariatric s | surgery within the | | | |
| <b>13</b> past 12 m | onths | S2085 PX | LAPAROSCOPIC GASTRIC BYPASS | CPT/HCPCS |
| Bariatric s | surgery within the | | LAPAROSCOPY, SURGICAL, GASTRIC RESTRICTIVE PROCEDURE; LONGITUDINAL | |
| 13 past 12 m | onths | 43775 PX | GASTRECTOMY (E.G., SLEEVE GASTRECTOMY) | CPT/HCPCS |
| Bariatric s | surgery within the | | | |
| 13 past 12 m | onths | 43848 PX | REVISION RYGB | CPT/HCPCS |


CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF


| Safety outcome: Urinary | | | |
|---|---|---|---|
| 7 tractinfection | CEFTAZIDIME IN DEXT RX | Generic | Urinary tract infection antibiotics |
| Safety outcome: Urinary<br>7 tract infection | CEFTAZIDIME SODIUM RX | Generic | Urinary tract infection antibiotics |
| Safety outcome: Urinary 7 tract infection | CEFTAZIDIME SODIUM RX | Generic | Urinary tract infection antibiotics |
| Safety outcome: Urinary 7 tract infection Safety outcome: Urinary | CEFTAZIDIME SODIUM RX | Generic | Urinary tract infection antibiotics |
| 7 tract infection<br>Safety outcome: Urinary | CEFTAZIDIME/ARGINITRX | Generic | Urinary tract infection antibiotics |
| 7 tract infection<br>Safety outcome: Urinary | CEFTAZIDIME/AVIBACRX | Generic | Urinary tract infection antibiotics |
| 7 tract infection<br>Safety outcome: Urinary | CEFTRIAXONE SODIUN RX | Generic | Urinary tract infection antibiotics |
| 7 tract infection<br>Safety outcome: Urinary | CEFTRIAXONE SODIUN RX | Generic | Urinary tract infection antibiotics |
| 7 tract infection<br>Safety outcome: Urinary | CEFTRIAXONE SODIUN RX | Generic | Urinary tract infection antibiotics |
| 7 tract infection<br>Safety outcome: Urinary | CEPHALEXIN RX | Generic | Urinary tract infection antibiotics |
| 7 tract infection<br>Safety outcome: Urinary | CEPHALEXIN HCL RX | Generic | Urinary tract infection antibiotics |
| 7 tract infection<br>Safety outcome: Urinary | CIPROFLOXACIN RX | Generic | Urinary tract infection antibiotics |
| 7 tract infection<br>Safety outcome: Urinary | CIPROFLOXACINHCL RX | Generic | Urinary tract infection antibiotics |
| 7 tract infection<br>Safety outcome: Urinary | CIPROFLOXACINLACTRX | Generic | Urinary tract infection antibiotics |
| 7 tract infection<br>Safety outcome: Urinary | CIPROFLOXACIN LAC1RX | Generic | Urinary tract infection antibiotics |
| 7 tract infection<br>Safety outcome: Urinary | CIPROFLOXACIN/CIPFRX | Generic | Urinary tract infection antibiotics |
| 7 tract infection<br>Safety outcome: Urinary | DORIPENEM RX | Generic | Urinary tract infection antibiotics |
| 7 tract infection<br>Safety outcome: Urinary | ERTAPENEM SODIUM RX | Generic | Urinary tract infection antibiotics |
| 7 tract infection<br>Safety outcome: Urinary | FOSFOMYCIN TROMET RX | Generic | Urinary tract infection antibiotics |
| 7 tract infection<br>Safety outcome: Urinary | GENTAMICIN SULFATERX | Generic | Urinary tract infection antibiotics |
| 7 tract infection<br>Safety outcome: Urinary | IMIPENEM/CILASTATII RX | Generic | Urinary tract infection antibiotics |
| 7 tract infection<br>Safety outcome: Urinary | IMIPENEM/CILASTATII RX | Generic | Urinary tract infection antibiotics |
| 7 tract infection<br>Safety outcome: Urinary | LEVOFLOXACIN RX | Generic | Urinary tract infection antibiotics |
| 7 tract infection<br>Safety outcome: Urinary | LEVOFLOXACIN/DEXT RX | Generic | Urinary tract infection antibiotics |
| 7 tract infection<br>Safety outcome: Urinary | MEROPENEM RX | Generic | Urinary tract infection antibiotics |
| 7 tract infection<br>Safety outcome: Urinary | MEROPENEM IN 0.9 % ! RX | Generic | Urinary tract infection antibiotics |
| 7 tract infection<br>Safety outcome: Urinary | MEROPENEM/VABORERX | Generic | Urinary tract infection antibiotics |
| 7 tract infection<br>Safety outcome: Urinary | NITROFURANTOIN RX | Generic | Urinary tract infection antibiotics |
| 7 tract infection<br>Safety outcome: Urinary | NITROFURANTOIN MAI RX | Generic | Urinary tract infection antibiotics |
| 7 tract infection<br>Safety outcome: Urinary | NITROFURANTOIN MOI RX | Generic | Urinary tract infection antibiotics |
| 7 tract infection<br>Safety outcome: Urinary | PIPERACILLIN AND TA RX | Generic | Urinary tract infection antibiotics |
| 7 tract infection<br>Safety outcome: Urinary | PIPERACILLIN SODIUN RX | Generic | Urinary tract infection antibiotics |
| 7 tractinfection | PIPERACILLIN SODIUN RX | Generic | Urinary tract infection antibiotics |


#### Appendix 3. Flowchart for cohort assembly

| OPTUM (May 13, 2022 to Feb 28, 2025) | | |
|---|---|---|
| | Excluded Patients | Remaining Patients |
| Patients in dataset | | 95,349,410 |
| Patients meeting cohort entry criteria | | 562,932 |
| Excluded due to insufficient enrollment | -206,396 (37%) | 356,536 |
| Excluded due to prior use of referent | -105,172 (29%) | 251,364 |
| Excluded due to prior use of exposure | -129,188 (51%) | 122,176 |
| Excluded because patient qualified in >1 exposure category | -3 (<1%) | 122,173 |
| Excluded based on 1 - Age | -29 (<1%) | 122,144 |
| Excluded based on 1 - Gender | -10 (<1%) | 122,134 |
| Excluded based on 2 - Type 2 diabetes mellitus | -5,202 (4%) | 116,932 |
| Excluded based on 3 - BMI ≥ 25kg/m2 (ICD-10) | -11,050 (9%) | 105,882 |
| Excluded based on 3 - BMI ≥ 25kg/m2 (Truncated) | -323 (<1%) | 105,559 |
| Excluded based on 4 - Increased cardiovascular risk | -1,562 (1%) | 103,997 |
| Excluded based on 5 - History of T1DM or secondary diabetes | -1,115 (1%) | 102,882 |
| Excluded based on 6 - Family or personal history of multiple endocrine neoplasia or medullary thyroid carcinoma | -171 (<1%) | 102,711 |
| Excluded based on 7 - End-stage renal disease or dialysis | -553 (<1%) | 102,158 |
| Excluded based on 8 - History of treatment for diabetic retinopathy and/or macular edema | -779 (<1%) | 101,379 |
| Excluded based on 9 - History of any malignancy | -3,124 (3%) | 98,255 |
| Excluded based on 10 - Cardiovascular event or intervention in the past 7 days | -45 (<1%) | 98,210 |
| Excluded based on 11 - Women who are pregnant or breastfeeding | -37 (<1%) | 98,173 |
| Excluded based on 12 - GLP-1-RA treatment within past 6 months | -5,422 (6%) | 92,751 |
| Excluded based on 13 - Bariatric surgery within the past 12 months | -233 (<1%) | 92,518 |
| Patients in Exposure Group | | 59,056 |
| Patients in Referent Group | | 33,462 |
| Total Patients | | 92,518 |

| MARKETSCAN (May 13, 2022 to Dec 31, 2023) | | |
|---|---|---|
| | Excluded Patients | Remaining Patients |
| Patients in dataset | | 126,118,01 |
| Patients meeting cohort entry criteria | | 319,215 |
| Excluded due to insufficient enrollment | -62,207 (19%) | 257,008 |
| Excluded due to prior use of referent | -96,869 (38%) | 160,139 |
| Excluded due to prior use of exposure | -90,744 (57%) | 69,395 |
| Excluded because patient qualified in >1 exposure category | -6 (<1%) | 69,389 |
| Excluded based on 1 - Age | -33 (<1%) | 69,356 |
| Excluded based on 1 - Gender | -0 (<1%) | 69,356 |
| Excluded based on 2 - Type 2 diabetes mellitus | -8,606 (12%) | 60,750 |
| Excluded based on 3 - BMI ≥ 25kg/m2 (ICD-10) | -7,643 (13%) | 53,107 |
| Excluded based on 4 - Increased cardiovascular risk | -1,638 (3%) | 51,469 |
| Excluded based on 5 - History of T1DM or secondary diabetes | -610 (1%) | 50,859 |
| Excluded based on 6 - Family or personal history of multiple endocrine neoplasia or medullary thyroid carcinoma | -110 (<1%) | 50,749 |
| Excluded based on 7 - End-stage renal disease or dialysis | -148 (<1%) | 50,60 |
| Excluded based on 8 - History of treatment for diabetic retinopathy and/or macular edema | -311 (<1%) | 50,290 |
| Excluded based on 9 - History of any malignancy | -1,371 (3%) | 48,919 |
| Excluded based on 10 - Cardiovascular event or intervention in the past 7 days | -33 (<1%) | 48,886 |
| Excluded based on 11 - Women who are pregnant or breastfeeding | -70 (<1%) | 48,816 |
| Excluded based on Censor: Other GLP-1-RA | -4,953 (10%) | 43,863 |
| Excluded based on 13 - Bariatric surgery within the past 12 months | -125 (<1%) | 43,738 |
| Patients in Exposure Group | | 23,797 |
| Patients in Referent Group | | 19,94 |
| Total Patients | | 43,738 |

#### Appendix 4.1st Feasibility Assessment

#### Table of Contents

- A. Patient characteristics by treatment group
- B. Summary Parameters of Study Population
- C. Median Follow up Time in Overall Study Population
- D. Reasons for Censoring in Overall Study Population
- E. Initial Power Assessment
- F. Aetion report link
- G. Review by Principal Investigator

In order to complete the initial power analysis, a dummy outcome of a 90-day gap in database enrollment was used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. We completed a PS overlap weighted comparative analysis using this outcome. The PS included only 3 covariates: age, sex, and combined comorbidity index. Power calculations are based on the formulas from Chow et al. (2008).

#### A. Patient characteristics by treatment group (follow-up start is 1 days after CED, so few patients and dropped, hence table 1 could include sightly fewer patients than the attrition table)

| Before matching | | Optum | | Marketscan | | |
|---|---|---|---|---|---|---|
| Variable | Reference: Dulaglutide | Exposure: Tirzepatide | Difference | Reference: Dulaglutide | Exposure: Tirzepatide | Difference |
| Number of patients | 33,462 | 59,056 | - (-, -) | 19,941 | 23,797 | - (-, -) |
| Age | | | | | | |
| mean (sd) | 64.56 (11.08) | 61.57 (11.51) | 2.99 (2.84, 3.14) | 56.41 (11.05) | 53.84 (10.02) | 2.58 (2.38, 2.78) |
| median [IQR] | 67.00 [58.00, 72.00] | 64.00 [54.00, 70.00] | - (-, -) | 57.00 [49.00, 63.00] | 54.00 [48.00, 60.00] | - (-, -) |
| Gender | | | | | | |
| Male; n (%) | 15,503 (46.3%) | 26,107 (44.2%) | 2.1% (1.5%, 2.8%) | 9,699 (48.6%) | 10,571 (44.4%) | 4.2% (3.3%, 5.2%) |
| CCI (365 days) | | | | | | |
| mean (sd) | 2.30 (2.61) | 1.80 (2.28) | 0.50 (0.47, 0.53) | 1.17 (1.81) | 0.93 (1.58) | 0.24 (0.21, 0.27) |
| median [IQR] | 2.00 [0.00, 4.00] | 1.00 [0.00, 3.00] | - (-, -) | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | - (-, -) |

#### B. Summary Parameters of Overall Study Population (Step 1)

| | Optum | Marketscan |
|-----------------------------------------------------|----------|-------------|
| Variable | Value | Value |
| Number of patients in full cohort | 92,518 | 43,738 |
| Number of patients dropped as incomplete cases | ( | 0 |
| Number of patients that did not begin follow-up | 143 | 3 |
| Number of patients in analytic cohort | 92,375 | 43,714 |
| Number of events | 1,02 | 236.00 |
| Number of person-years | 46,911.7 | 1 20,227.33 |
| Number of patients in group: Reference-Sitagliptin | 33,420 | 19,927 |
| Number of patients in group: Exposure - Tirzepatide | 58,955 | 23,787 |
| Risk per 1,000 patients | 11.06 | 5.4 |
| Rate per 1,000 person-years | 21.79 | 11.67 |

#### C. Median Follow up Time in Overall Study Population (Step 1)

| | Optum | Marketscan |
|----------------------------|------------------|------------------|
| Patient Group | Median Follow-Up | Median Follow-Up |
| Overall Patient Population | 154 [74, 299] | 143 [71, 256] |

#### D. Reasons for Censoring in Overall Study Population (Step 1)

| Optum | Marketscan |
|-------|------------|

| Overall | Value | Value |
|---|---|---|
| Outcome | 1,022 (1.1%) | 236 (0.5%) |
| Start of an additional exposure | 1,958 (2.1%) | 1,122 (2.6%) |
| End of index exposure | 36,034 (39.0%) | 11,304 (25.9%) |
| Maximum follow-up time | 16,860 (18.3%) | 4,703 (10.8%) |
| Specified date reached | 6,999 (7.6%) | 21,493 (49.2%) |
| End of patient data | 0 (0.0%) | 0 (0.0%) |
| End of patient enrollment | 24,018 (26.0%) | 3,049 (7.0%) |
| Switch to other GLP-1-RA (for censoring) / Nursing home admission | 5,484 (5.9%) | 1,807 (4.1%) |

#### E. Power Assessment

| Noninferiority Analysis | Optum | Marketscan |
|----------------------------|--------|------------|
| Number of patients matched | | |
| Reference | 33,462 | 19,941 |
| Exposed | 59,056 | 23,797 |
| Risk per 1,000 patients | 11.06 | 5.4 |
| Assumed HR from RCT | 0.8 | 0.8 |
| Alpha (2-sided) | 0.05 | 0.05 |
| Non-inferiority margin | 1.05 | 1.05 |
| Number of events expected | 1023 | 236 |
| Power | 0.99 | 0.55 |

## F. Aetion report link

Optum Step 1: https://bwh-dopeaetion.com/project/2905/rwrs/139333

Marketscan Step 1: https://bwh-dopeaetion.com/project/2906/rwrs/139337

## F. Review by principal investigator

Stop analyses until feasibility and power are reviewed by primary investigators.

| Reviewed by PI: | Nils Krüger | Date reviewed: | July 30, 2025 |
|-----------------|-------------|----------------|---------------|

## Appendix 5. 2nd Feasibility Assessment

## **Table of Contents**

A. Median Follow up Time by Treatment Group

B. Reasons for Censoring by Treatment Group

C. Final Power Assessment

D. Aetion report link

E. Review by Principal Investigator

In order to complete the feasibility analysis, a dummy outcome of a 90-day gap in database enrollment was used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. We completed a PS overlap weighted comparative analysis using this outcome. The PS included all prespecified covariates listed in the protocol. Power calculations are based on the formulas from Chow et al. (2008).

# A. Median Follow Up Time by Treatment Group

| | Median Follow-Up | Median Follow-Up |
|----------------------------|-------------------|-------------------|
| Patient Group | Time (Days) [IQR] | Time (Days) [IQR] |
| Overall Patient Population | 154 [74, 299] | 143 [71, 256] |

# **B.** Reasons for Censoring in Overall Study Population

| | Optum | Marketscan |
|---|---|---|
| Overall | Value | Value |
| Outcome | 1,022 (1.1%) | 236 (0.5%) |
| Start of an additional exposure | 1,958 (2.1%) | 1,122 (2.6%) |
| End of index exposure | 36,034 (39.0%) | 11,304 (25.9%) |
| Maximum follow-up time | 16,860 (18.3%) | 4,703 (10.8%) |
| Specified date reached | 6,999 (7.6%) | 21,493 (49.2%) |
| End of patient data | 0 (0.0%) | 0 (0.0%) |
| End of patient enrollment | 24,018 (26.0%) | 3,049 (7.0%) |
| Switch to other GLP-1-RA (for censoring) / Nursing home admission | 5,484 (5.9%) | 1,807 (4.1%) |

## **C. Power Assessment**

| Noninferiority Analysis | Optum | Marketscan |
|----------------------------|-------|------------|
| Number of patients matched | | |

| Reference | 33,462 | 19,941 |
|---------------------------|--------|--------|
| Exposed | 59,056 | 23,797 |
| Risk per 1,000 patients | 11.06 | 5.4 |
| Assumed HR from RCT | 0.8 | 0.8 |
| Alpha (2-sided) | 0.05 | 0.05 |
| Non-inferiority margin | 1.05 | 1.05 |
| Number of events expected | 1023 | 236 |
| Power | 0.99 | 0.55 |

# D. Aetion report link

Optum Step 1: https://bwh-dope.aetion.com/project/2905/rwrs/139333
Marketscan Step 1: https://bwh-dope.aetion.com/project/2906/rwrs/139337

## E. Review by principal investigator

Stop analyses until feasibility and power are reviewed by primary investigators.

| Reviewed by PI: | Nils Krüger | Date reviewed: | July 30, 2025 |
|-----------------|-------------|----------------|---------------|
|-----------------|-------------|----------------|---------------|

## Appendix 6. Balance Assessment - PS Distribution and C-Statistic

C-statistics unadjusted, OPTUM: 0.772



C-statistics adjusted after overlap weighing on the PS, OPTUM: 0.514



C-statistics unadjusted, MARKETSCAN: 0.721



C-statistics adjusted after overlap weighing on the PS, MARKETSCAN: 0.521



Appendix 7. Balance Assessment - Table 1

| | 1 | | | | | |
|---|---|---|---|---|---|---|
| OPTUM | | | | | | |
| Variable | Reference: Dulaglutide | Exposure: Tirzepatide | Difference | Reference: Dulaglutide | Exposure: Tirzepatide | Difference |
| Number of patients | 33,420 | 58,955 | - (-, -) | 24,795 | 24,795 | - (-, -) |
| Year of Cohort Entry Date | | | | | | |
| 2022; n (%) | 11,086 (33.2%) | 5,070 (8.6%) | 24.6% (24.0%, 25.1%) | 4,679 (18.9%) | 4,714 (19.0%) | -0.1% (-0.8%, 0.6%) |
| 2023; n (%) | 14,561 (43.6%) | 23,677 (40.2%) | 3.4% (2.7%, 4.1%) | 12,554 (50.6%) | 12,453 (50.2%) | 0.4% (-0.5%, 1.3%) |
| 2024; n (%) | 7,632 (22.8%) | 28,830 (48.9%) | -26.1% (-26.7%, -25.5%) | 7,421 (29.9%) | 7,487 (30.2%) | -0.3% (-1.1%, 0.5%) |
| 2025; n (%) | 141 (0.4%) | 1,378 (2.3%) | -1.9% (-2.1%, -1.8%) | 141 (0.6%) | 141 (0.6%) | 0.0% (-0.1%, 0.1%) |
| Age | | | | | | |
| mean (sd) | 64.56 (11.07) | 61.57 (11.51) | 2.99 (2.84, 3.15) | 63.46 (11.20) | 63.44 (11.03) | 0.02 (-0.18, 0.22) |
| median [IQR] | 67.00 [58.00, 72.00] | 64.00 [54.00, 70.00] | - (-, -) | 66.00 [56.00, 71.00] | 66.00 [56.00, 71.00] | - (-, -) |
| min, max | 18.00, 88.00 | 18.00, 88.00 | - (-, -) | 18.00, 88.00 | 18.00, 88.00 | - (-, -) |
| Gender (male); n (%) | 15,486 (46.3%) | 26,058 (44.2%) | 2.1% (1.5%, 2.8%) | 11,312 (45.6%) | 11,294 (45.5%) | 0.1% (-0.8%, 1.0%) |
| Race (Recategorized) | | | | | | |
| .White: n (%) | 14.596 (43.7%) | 26.911 (45.6%) | -2.0% (-2.6%, -1.3%) | 10.965 (44.2%) | 10.963 (44.2%) | 0.0% (-0.9%, 0.9%) |
| .Black: n (%) | 4.928 (14.7%) | 7.226 (12.3%) | 2.5% (2.0%, 3.0%) | 3.449 (13.9%) | 3,480 (14,0%) | -0.1% (-0.7%, 0.5%) |
| .Unknown / Missing; n (%) | 13,350 (39.9%) | 23,995 (40.7%) | -0.8% (-1.4%, -0.1%) | 10,009 (40.4%) | 9,964 (40.2%) | 0.2% (-0.7%, 1.0%) |
| Others; n (%) | 546 (1.6%) | 823 (1.4%) | 0.2% (0.1%, 0.4%) | 372 (1.5%) | 388 (1.6%) | -0.1% (-0.3%, 0.2%) |
| Region / State | 370 (1.070) | OLO (1.770) | 5.E/6 (5.1/6, 5.T/0) | 3,2(13/0) | 000 (1.070) | J.170 ( J.J 70, U.Z 70) |
| Northest; n (%) | 3,469 (10.4%) | 4,411 (7.5%) | 2.9% (2.5%, 3.3%) | 2,226 (9.0%) | 2,214 (8.9%) | 0.0% (-0.5%, 0.6%) |
| | 7,692 (23.0%) | 12,719 (21.6%) | 1.4% (0.9%, 2.0%) | 5,735 (23.1%) | 5,719 (23.1%) | 0.0% (-0.5%, 0.6%) |
| .Midwest / North central; n (%) | | T . | | | | |
| South; n (%) | 15,773 (47.2%) | 34,090 (57.8%) | -10.6% (-11.3%, -10.0%) | 12,534 (50.6%) | 12,586 (50.8%) | -0.2% (-1.1%, 0.7%) |
| .West; n (%) | 6,473 (19.4%) | 7,700 (13.1%) | 6.3% (5.8%, 6.8%) | 4,289 (17.3%) | 4,268 (17.2%) | 0.1% (-0.6%, 0.8%) |
| .Missing; n (%) | 13 (0.0%) | 35 (0.1%) | -0.0% (-0.1%, 0.0%) | 11 (0.0%) | 8 (0.0%) | 0.0% (-0.0%, 0.1%) |
| Smoking/Tobacco use; n (%) | 8,434 (25.2%) | 13,408 (22.7%) | 2.5% (1.9%, 3.1%) | 6,038 (24.4%) | 6,002 (24.2%) | 0.1% (-0.6%, 0.9%) |
| Veight | | | | | | |
| Overweight; n (%) | 3,734 (11.2%) | 3,573 (6.1%) | 5.1% (4.7%, 5.5%) | 2,219 (8.9%) | 2,244 (9.1%) | -0.1% (-0.6%, 0.4%) |
| .Class 1 Obesity; n (%) | 7,515 (22.5%) | 10,345 (17.5%) | 4.9% (4.4%, 5.5%) | 5,161 (20.8%) | 5,144 (20.7%) | 0.1% (-0.6%, 0.8%) |
| .Class 2 Obesity; n (%) | 9,753 (29.2%) | 18,370 (31.2%) | -2.0% (-2.6%, -1.4%) | 7,502 (30.3%) | 7,578 (30.6%) | -0.3% (-1.1%, 0.5%) |
| .Class 3 Obesity; n (%) | 7,889 (23.6%) | 18,355 (31.1%) | -7.5% (-8.1%, -6.9%) | 6,469 (26.1%) | 6,455 (26.0%) | 0.1% (-0.7%, 0.8%) |
| .Unspecified Obesity; n (%) | 4,529 (13.6%) | 8,312 (14.1%) | -0.5% (-1.0%, -0.1%) | 3,444 (13.9%) | 3,374 (13.6%) | 0.3% (-0.3%, 0.9%) |
| Diabetic retinopathy; n (%) | 4,065 (12.2%) | 4,491 (7.6%) | 4.5% (4.1%, 5.0%) | 2,605 (10.5%) | 2,576 (10.4%) | 0.1% (-0.4%, 0.7%) |
| Diabetic neuropathy; n (%) | 11,222 (33.6%) | 13,958 (23.7%) | 9.9% (9.3%, 10.5%) | 7,468 (30.1%) | 7,516 (30.3%) | -0.2% (-1.0%, 0.6%) |
| Diabetic nephropathy; n (%) | 9,023 (27.0%) | 11,313 (19.2%) | 7.8% (7.2%, 8.4%) | 5,981 (24.1%) | 6,027 (24.3%) | -0.2% (-0.9%, 0.6%) |
| Diabetes with other ophthalmic complications; n (%) | 1,798 (5.4%) | 2,082 (3.5%) | 1.8% (1.6%, 2.1%) | 1,149 (4.6%) | 1,159 (4.7%) | -0.0% (-0.4%, 0.3%) |
| Diabetes with peripheral circulatory disorders; n (%) | 5,992 (17.9%) | 7,667 (13.0%) | 4.9% (4.4%, 5.4%) | 3,957 (16.0%) | 3,968 (16.0%) | -0.0% (-0.7%, 0.6%) |
| Diabetic foot; n (%) | 1,358 (4.1%) | 1,608 (2.7%) | 1.3% (1.1%, 1.6%) | 860 (3.5%) | 877 (3.5%) | -0.1% (-0.4%, 0.3%) |
| rectile dysfunction; n (%) | 1,708 (5.1%) | 2,918 (4.9%) | 0.2% (-0.1%, 0.5%) | 1,259 (5.1%) | 1,253 (5.1%) | 0.0% (-0.4%, 0.4%) |
| Typoglycemia; n (%) | 9,056 (27.1%) | 14,423 (24.5%) | 2.6% (2.0%, 3.2%) | 6,416 (25.9%) | 6,481 (26.1%) | -0.3% (-1.0%, 0.5%) |
| Typerglycemia/DKA/HONK; n (%) | 19,342 (57.9%) | 29,255 (49.6%) | 8.3% (7.6%, 8.9%) | 13,634 (55.0%) | 13,717 (55.3%) | -0.3% (-1.2%, 0.5%) |
| Skin infections; n (%) | 3,863 (11.6%) | 6,255 (10.6%) | 0.9% (0.5%, 1.4%) | 2,739 (11.0%) | 2,735 (11.0%) | 0.0% (-0.5%, 0.6%) |
| stable angina; n (%) | 1,664 (5.0%) | 2,540 (4.3%) | 0.7% (0.4%, 1.0%) | 1,168 (4.7%) | 1,191 (4.8%) | -0.1% (-0.5%, 0.3%) |
| Instable angina; n (%) | 883 (2.6%) | 1.301 (2.2%) | 0.4% (0.2%, 0.6%) | 615 (2.5%) | 640 (2.6%) | -0.1% (-0.4%, 0.2%) |
| Instable angina; n (%) Ivpertension: n (%) | 29.914 (89.5%) | 1,301 (2.2%)<br>51.511 (87.4%) | 2.1% (1.7%, 2.6%) | 22.005 (88.7%) | 21,980 (88.6%) | 0.1% (-0.5%, 0.7%) |
| 77 | 1,290 (3.9%) | 1,621 (2.7%) | 2.1% (1.7%, 2.6%)<br>1.1% (0.9%, 1.4%) | 812 (3.3%) | 21,980 (88.6%)<br>807 (3.3%) | 0.1% (-0.5%, 0.7%) |
| Hypotension; n (%) | | | | | | |
| Hyperlipidemia; n (%) | 28,764 (86.1%) | 49,978 (84.8%) | 1.3% (0.8%, 1.8%) | 21,210 (85.5%) | 21,234 (85.6%) | -0.1% (-0.7%, 0.5%) |
| Atrial fibrillation; n (%) | 3,542 (10.6%) | 5,456 (9.3%) | 1.3% (0.9%, 1.8%) | 2,416 (9.7%) | 2,412 (9.7%) | 0.0% (-0.5%, 0.5%) |
| Cardiac conduction disorder; n (%) | 2,179 (6.5%) | 3,130 (5.3%) | 1.2% (0.9%, 1.5%) | 1,458 (5.9%) | 1,440 (5.8%) | 0.1% (-0.3%, 0.5%) |
| Previous cardiac procedure (CABG, PTCA, Stent); n (%) | 577 (1.7%) | 772 (1.3%) | 0.4% (0.2%, 0.6%) | 379 (1.5%) | 389 (1.6%) | -0.0% (-0.3%, 0.2% |
| schemic stroke; n (%) | 316 (0.9%) | 284 (0.5%) | 0.5% (0.3%, 0.6%) | 171 (0.7%) | 169 (0.7%) | 0.0% (-0.1%, 0.2%) |
| VD diagnosis or surgery; n (%) | 3,923 (11.7%) | 4,970 (8.4%) | 3.3% (2.9%, 3.7%) | 2,551 (10.3%) | 2,574 (10.4%) | -0.1% (-0.6%, 0.4%) |
| ther cardiac dysrhythmia; n (%) | 6,939 (20.8%) | 11,624 (19.7%) | 1.0% (0.5%, 1.6%) | 4,932 (19.9%) | 4,919 (19.8%) | 0.1% (-0.7%, 0.8%) |
| ardiomyopathy; n (%) | 1,930 (5.8%) | 2,644 (4.5%) | 1.3% (1.0%, 1.6%) | 1,270 (5.1%) | 1,286 (5.2%) | -0.1% (-0.5%, 0.3%) |
| /alve disorders; n (%) | 3,785 (11.3%) | 5,942 (10.1%) | 1.2% (0.8%, 1.7%) | 2,635 (10.6%) | 2,627 (10.6%) | 0.0% (-0.5%, 0.6%) |
| /alve replacement; n (%) | 398 (1.2%) | 608 (1.0%) | 0.2% (0.0%, 0.3%) | 282 (1.1%) | 298 (1.2%) | -0.1% (-0.3%, 0.1%) |
| TA; n (%) | 681 (2.0%) | 876 (1.5%) | 0.6% (0.4%, 0.7%) | 440 (1.8%) | 411 (1.7%) | 0.1% (-0.1%, 0.3%) |
| Edema; n (%) | 4,894 (14.6%) | 8,052 (13.7%) | 1.0% (0.5%, 1.5%) | 3,450 (13.9%) | 3,440 (13.9%) | 0.0% (-0.6%, 0.7%) |
| /enous thromboembolism / Pulmonary embolism; n (%) | 1,226 (3.7%) | 1,880 (3.2%) | 0.5% (0.2%, 0.7%) | 807 (3.3%) | 818 (3.3%) | -0.0% (-0.4%, 0.3% |
| Pulmonary hypertension; n (%) | 1,081 (3.2%) | 1,689 (2.9%) | 0.4% (0.1%, 0.6%) | 749 (3.0%) | 744 (3.0%) | 0.0% (-0.3%, 0.3%) |
| mplantable cardioverter defibrillator; n (%) | 105 (0.3%) | 142 (0.2%) | 0.1% (-0.0%, 0.1%) | 78 (0.3%) | 72 (0.3%) | 0.0% (-0.1%, 0.1%) |
| inplantable caraloverter defibrillator, 11 (70) | 100 (0.070) | 172 (0.2/0) | U.170 (-U.U /U, U.170) | 10 (0.070) | 12 (0.0 /0) | 0.070 (-0.170, 0.170) |

| Hyperkalemia; n (%) | 1,379 (4.1%) | 1,476 (2.5%) | 1.6% (1.4%, 1.9%) | 803 (3.2%) | 835 (3.4%) | -0.1% (-0.4%, 0.2%) |
|---|---|---|---|---|---|---|
| Coronary atherosclerosis: n (%) | 7.770 (23.2%) | 11.680 (19.8%) | 3.4% (2.9%, 4.0%) | 5.428 (21.9%) | 5.497 (22.2%) | -0.3% (-1.0%, 0.5%) |
| Cerebrovascular procedure; n (%) | 55 (0.2%) | 53 (0.1%) | 0.1% (0.0%, 0.1%) | 29 (0.1%) | 31 (0.1%) | -0.0% (-0.1%, 0.1%) |
| Insertion of pacemakers / removal of cardiac lead; n (%) | 68 (0.2%) | 89 (0.2%) | 0.1% (-0.0%, 0.1%) | 45 (0.2%) | 44 (0.2%) | 0.0% (-0.1%, 0.1%) |
| CKD Stage 1-2; n (%) | 2,026 (6.1%) | 2,919 (5.0%) | 1.1% (0.8%, 1.4%) | 1,404 (5.7%) | 1,401 (5.7%) | 0.0% (-0.4%, 0.4%) |
| CKD Stage 3-4; n (%) | 6,530 (19.5%) | 8,085 (13.7%) | 5.8% (5.3%, 6.3%) | 4,283 (17.3%) | 4,316 (17.4%) | -0.1% (-0.8%, 0.5%) |
| Unspecified CKD; n (%) | 2,641 (7.9%) | 3,084 (5.2%) | 2.7% (2.3%, 3.0%) | 1,634 (6.6%) | 1,672 (6.7%) | -0.2% (-0.6%, 0.3%) |
| Acute kidney injury; n (%) | 2,810 (8.4%) | 3,067 (5.2%) | 3.2% (2.9%, 3.6%) | 1,702 (6.9%) | 1,699 (6.9%) | 0.0% (-0.4%, 0.5%) |
| Hypertensive nephropathy; n (%) | 5,451 (16.3%) | 6,647 (11.3%) | 5.0% (4.6%, 5.5%) | 3,519 (14.2%) | 3,530 (14.2%) | -0.0% (-0.7%, 0.6%) |
| Urinary tract infections; n (%) | 4,841 (14.5%) | 7,575 (12.8%) | 1.6% (1.2%, 2.1%) | 3,344 (13.5%) | 3,353 (13.5%) | -0.0% (-0.6%, 0.6%) |
| Genital infections; n (%) | 1,217 (3.6%) | 1,632 (2.8%) | 0.9% (0.6%, 1.1%) | 776 (3.1%) | 813 (3.3%) | -0.1% (-0.5%, 0.2%) |
| Urolithiasis (Kidney and urinary stone); n (%) | 1,480 (4.4%) | 2,751 (4.7%) | -0.2% (-0.5%, 0.0%) | 1,116 (4.5%) | 1,080 (4.4%) | 0.1% (-0.2%, 0.5%) |
| COPD; n (%) | 4,782 (14.3%) | 6,763 (11.5%) | 2.8% (2.4%, 3.3%) | 3,258 (13.1%) | 3,260 (13.1%) | -0.0% (-0.6%, 0.6%) |
| Asthma; n (%) | 3,955 (11.8%) | 7,580 (12.9%) | -1.0% (-1.5%, -0.6%) | 3,010 (12.1%) | 3,027 (12.2%) | -0.1% (-0.6%, 0.5%) |
| Obstructive sleep apnea; n (%) | 9,689 (29.0%) | 20,297 (34.4%) | -5.4% (-6.1%, -4.8%) | 7,585 (30.6%) | 7,681 (31.0%) | -0.4% (-1.2%, 0.4%) |
| Serious bacterial infections; n (%) | 1,244 (3.7%) | 1,435 (2.4%) | 1.3% (1.0%, 1.5%) | 751 (3.0%) | 726 (2.9%) | 0.1% (-0.2%, 0.4%) |
| Pneumonia; n (%) | 1,858 (5.6%) | 2,449 (4.2%) | 1.4% (1.1%, 1.7%) | 1,162 (4.7%) | 1,149 (4.6%) | 0.1% (-0.3%, 0.4%) |
| Liver disease; n (%) | 5,938 (17.8%) | 10,714 (18.2%) | -0.4% (-0.9%, 0.1%) | 4,371 (17.6%) | 4,446 (17.9%) | -0.3% (-1.0%, 0.4%) |
| MASH/MASLD; n (%) | 3,047 (9.1%) | 6,574 (11.2%) | -2.0% (-2.4%, -1.6%) | 2,435 (9.8%) | 2,439 (9.8%) | -0.0% (-0.5%, 0.5%) |
| Fractures / Falls; n (%) | 2,422 (7.2%) | 3,277 (5.6%) | 1.7% (1.4%, 2.0%) | 1,553 (6.3%) | 1,589 (6.4%) | -0.1% (-0.6%, 0.3%) |
| Osteoporosis; n (%) | 1,545 (4.6%) | 2,352 (4.0%) | 0.6% (0.4%, 0.9%) | 1,079 (4.4%) | 1,065 (4.3%) | 0.1% (-0.3%, 0.4%) |
| Osteoarthritis; n (%) | 10,341 (30.9%) | 17,956 (30.5%) | 0.5% (-0.1%, 1.1%) | 7,609 (30.7%) | 7,565 (30.5%) | 0.2% (-0.6%, 1.0%) |
| Depression; n (%) | 7,747 (23.2%) | 12,691 (21.5%) | 1.7% (1.1%, 2.2%) | 5,481 (22.1%) | 5,522 (22.3%) | -0.2% (-0.9%, 0.6%) |
| Dementia; n (%) | 1,775 (5.3%) | 1,475 (2.5%) | 2.8% (2.5%, 3.1%) | 904 (3.6%) | 917 (3.7%) | -0.1% (-0.4%, 0.3%) |
| Delirium or psychosis; n (%) | 859 (2.6%) | 767 (1.3%) | 1.3% (1.1%, 1.5%) | 458 (1.8%) | 462 (1.9%) | -0.0% (-0.3%, 0.2%) |
| Anxiety; n (%) | 7,344 (22.0%) | 14,178 (24.0%) | -2.1% (-2.6%, -1.5%) | 5,505 (22.2%) | 5,543 (22.4%) | -0.2% (-0.9%, 0.6%) |
| Sleep disorders; n (%) | 11,586 (34.7%) | 21,114 (35.8%) | -1.1% (-1.8%, -0.5%) | 8,576 (34.6%) | 8,579 (34.6%) | -0.0% (-0.9%, 0.8%) |
| Anemia; n (%) | 6,622 (19.8%) | 10,461 (17.7%) | 2.1% (1.5%, 2.6%) | 4,555 (18.4%) | 4,620 (18.6%) | -0.3% (-0.9%, 0.4%) |
| Influenza; n (%) | 567 (1.7%) | 1,283 (2.2%) | -0.5% (-0.7%, -0.3%) | 450 (1.8%) | 455 (1.8%) | -0.0% (-0.3%, 0.2%) |
| COVID; n (%) | 3,995 (12.0%) | 6,286 (10.7%) | 1.3% (0.9%, 1.7%) | 2,765 (11.2%) | 2,798 (11.3%) | -0.1% (-0.7%, 0.4%) |
| Hyperthyroidism and other thyroid gland disorders; n (%) | 8,261 (24.7%) | 15,598 (26.5%) | -1.7% (-2.3%, -1.2%) | 6,177 (24.9%) | 6,285 (25.3%) | -0.4% (-1.2%, 0.3%) |
| Hypothyroidism; n (%) | 6,685 (20.0%) | 12,630 (21.4%) | -1.4% (-2.0%, -0.9%) | 5,006 (20.2%) | 5,079 (20.5%) | -0.3% (-1.0%, 0.4%) |
| Nephrotic syndrome; n (%) | 43 (0.1%) | 46 (0.1%) | 0.1% (0.0%, 0.1%) | 27 (0.1%) | 23 (0.1%) | 0.0% (-0.0%, 0.1%) |
| Urinary incontinence; n (%) | 2,132 (6.4%) | 3,185 (5.4%) | 1.0% (0.7%, 1.3%) | 1,439 (5.8%) | 1,462 (5.9%) | -0.1% (-0.5%, 0.3%) |
| Biliary disease; n (%) | 70 (0.2%) | 68 (0.1%) | 0.1% (0.0%, 0.2%) | 42 (0.2%) | 44 (0.2%) | -0.0% (-0.1%, 0.1%) |
| Pancreatitis; n (%) | 38 (0.1%) | 57 (0.1%) | 0.0% (-0.0%, 0.1%) | 31 (0.1%) | 26 (0.1%) | 0.0% (-0.0%, 0.1%) |
| Bowel obstruction; n (%) | 44 (0.1%) | 76 (0.1%) | 0.0% (-0.0%, 0.1%) | 29 (0.1%) | 28 (0.1%) | 0.0% (-0.1%, 0.1%) |
| Gastroparesis; n (%) | 333 (1.0%) | 541 (0.9%) | 0.1% (-0.1%, 0.2%) | 250 (1.0%) | 254 (1.0%) | -0.0% (-0.2%, 0.2%) |
| Number of antidiabetic drugs on CED | | | | | | |
| mean (sd) | 2.36 (1.00) | 2.08 (0.96) | 0.28 (0.27, 0.29) | 2.27 (0.97) | 2.28 (1.02) | -0.01 (-0.03, 0.01) |
| median [IQR] | 2.00 [2.00, 3.00] | 2.00 [1.00, 3.00] | - (-, -) | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | - (-, -) |
| min, max | 1.00, 7.00 | 1.00, 7.00 | - (-, -) | 1.00, 7.00 | 1.00, 7.00 | - (-, -) |
| Concomitant use or initiation of Metformin; n (%) | 17,289 (51.7%) | 28,425 (48.2%) | 3.5% (2.8%, 4.2%) | 12,731 (51.3%) | 12,756 (51.4%) | -0.1% (-1.0%, 0.8%) |
| Concomitant use or initiation of Insulins; n (%) | 8,833 (26.4%) | 10,264 (17.4%) | 9.0% (8.5%, 9.6%) | 5,740 (23.1%) | 5,811 (23.4%) | -0.3% (-1.0%, 0.5%) |
| Concomitant use or initiation of Sulfonylureas; n (%) | 7,454 (22.3%) | 8,369 (14.2%) | 8.1% (7.6%, 8.6%) | 4,853 (19.6%) | 4,859 (19.6%) | -0.0% (-0.7%, 0.7%) |
| Concomitant use or initiation of DPP-4i; n (%) | 2,479 (7.4%) | 3,087 (5.2%) | 2.2% (1.8%, 2.5%) | 1,564 (6.3%) | 1,639 (6.6%) | -0.3% (-0.7%, 0.1%) |
| Concomitant use or initiation of SGLT-2i; n (%) | 6,928 (20.7%) | 10,133 (17.2%) | 3.5% (3.0%, 4.1%) | 4,962 (20.0%) | 4,996 (20.1%) | -0.1% (-0.8%, 0.6%) |
| Concomitant use or initiation of Any other glucose-lowering drugs; n (%) | 2,338 (7.0%) | 3,268 (5.5%) | 1.5% (1.1%, 1.8%) | 1,657 (6.7%) | 1,673 (6.7%) | -0.1% (-0.5%, 0.4%) |
| Past use of Metformin; n (%) | 22,648 (67.8%) | 37,945 (64.4%) | 3.4% (2.8%, 4.0%) | 16,705 (67.4%) | 16,764 (67.6%) | -0.2% (-1.1%, 0.6%) |
| Past use of Insulins; n (%) | 11,589 (34.7%) | 13,583 (23.0%) | 11.6% (11.0%, 12.3%) | 7,608 (30.7%) | 7,691 (31.0%) | -0.3% (-1.2%, 0.5%) |
| Past use of Sulfonylureas; n (%) | 10,386 (31.1%) | 12,080 (20.5%) | 10.6% (10.0%, 11.2%) | 6,872 (27.7%) | 6,911 (27.9%) | -0.2% (-0.9%, 0.6%) |
| Past use of DPP-4i; n (%) | 3,985 (11.9%) | 4,981 (8.4%) | 3.5% (3.1%, 3.9%) | 2,564 (10.3%) | 2,644 (10.7%) | -0.3% (-0.9%, 0.2%) |
| Past use of SGLT-2i; n (%) | 9,538 (28.5%) | 14,104 (23.9%) | 4.6% (4.0%, 5.2%) | 6,867 (27.7%) | 6,890 (27.8%) | -0.1% (-0.9%, 0.7%) |
| Past use of Any other glucose-lowering drugs; n (%) | 3,363 (10.1%) | 4,578 (7.8%) | 2.3% (1.9%, 2.7%) | 2,337 (9.4%) | 2,385 (9.6%) | -0.2% (-0.7%, 0.3%) |
| ACE-is/ARB's; n (%) | 25,033 (74.9%) | 42,276 (71.7%) | 3.2% (2.6%, 3.8%) | 18,365 (74.1%) | 18,387 (74.2%) | -0.1% (-0.9%, 0.7%) |
| ARNI; n (%) | 605 (1.8%) | 1,021 (1.7%) | 0.1% (-0.1%, 0.3%) | 447 (1.8%) | 450 (1.8%) | -0.0% (-0.3%, 0.2%) |
| Thiazides; n (%) | 11,075 (33.1%) | 20,857 (35.4%) | -2.2% (-2.9%, -1.6%) | 8,388 (33.8%) | 8,420 (34.0%) | -0.1% (-1.0%, 0.7%) |
| Beta-blockers; n (%) | 14,764 (44.2%) | 23,685 (40.2%) | 4.0% (3.3%, 4.7%) | 10,535 (42.5%) | 10,517 (42.4%) | 0.1% (-0.8%, 0.9%) |
| Calcium channel blockers; n (%) | 11,543 (34.5%) | 18,824 (31.9%) | 2.6% (2.0%, 3.2%) | 8,286 (33.4%) | 8,352 (33.7%) | -0.3% (-1.1%, 0.6%) |
| Digoxin / Digitoxin; n (%) | 248 (0.7%) | 300 (0.5%) | 0.2% (0.1%, 0.3%) | 157 (0.6%) | 149 (0.6%) | 0.0% (-0.1%, 0.2%) |
| Loop diuretics; n (%) | 6,693 (20.0%) | 10,407 (17.7%) | 2.4% (1.8%, 2.9%) | 4,678 (18.9%) | 4,743 (19.1%) | -0.3% (-1.0%, 0.4%) |
| Other diuretics; n (%) | 3,042 (9.1%) | 5,445 (9.2%) | -0.1% (-0.5%, 0.3%) | 2,270 (9.2%) | 2,321 (9.4%) | -0.2% (-0.7%, 0.3%) |

| Intravenous diuretics; n (%) | 545 (1.6%) | 746 (1.3%) | 0.4% (0.2%, 0.5%) | 347 (1.4%) | 359 (1.4%) | -0.0% (-0.3%, 0.2%) |
|---|---|---|---|---|---|---|
| Nitrates; n (%) | 2,469 (7.4%) | 3,331 (5.7%) | 1.7% (1.4%, 2.1%) | 1,678 (6.8%) | 1,732 (7.0%) | -0.2% (-0.7%, 0.2%) |
| Anti-arrhythmics; n (%) | 722 (2.2%) | 1,351 (2.3%) | -0.1% (-0.3%, 0.1%) | 538 (2.2%) | 529 (2.1%) | 0.0% (-0.2%, 0.3%) |
| Statins; n (%) | 28,084 (84.0%) | 45,331 (76.9%) | 7.1% (6.6%, 7.7%) | 20,433 (82.4%) | 20,415 (82.3%) | 0.1% (-0.6%, 0.7%) |
| PCSK9 inhibitors and other lipid-lowering drugs; n (%) | 4,452 (13.3%) | 8,255 (14.0%) | -0.7% (-1.1%, -0.2%) | 3,410 (13.8%) | 3,428 (13.8%) | -0.1% (-0.7%, 0.5%) |
| Antiplatelet medications; n (%) | 3,755 (11.2%) | 5,279 (9.0%) | 2.3% (1.9%, 2.7%) | 2,555 (10.3%) | 2,574 (10.4%) | -0.1% (-0.6%, 0.5%) |
| Oral anticoagulants; n (%) | 3,805 (11.4%) | 5,812 (9.9%) | 1.5% (1.1%, 1.9%) | 2,609 (10.5%) | 2,618 (10.6%) | -0.0% (-0.6%, 0.5%) |
| COPD/Asthma medications; n (%) | 11,741 (35.1%) | 21,806 (37.0%) | -1.9% (-2.5%, -1.2%) | 8,851 (35.7%) | 8,840 (35.7%) | 0.0% (-0.8%, 0.9%) |
| NSAIDS; n (%) | 10,685 (32.0%) | 19,911 (33.8%) | -1.8% (-2.4%, -1.2%) | 8,051 (32.5%) | 8,030 (32.4%) | 0.1% (-0.7%, 0.9%) |
| Oral corticosteroids; n (%) | 7,323 (21.9%) | 16,517 (28.0%) | -6.1% (-6.7%, -5.5%) | 5,875 (23.7%) | 5,873 (23.7%) | 0.0% (-0.7%, 0.8%) |
| Osteoporosis agents (incl. bisphosphonates); n (%) | 959 (2.9%) | 1,380 (2.3%) | 0.5% (0.3%, 0.7%) | 676 (2.7%) | 666 (2.7%) | 0.0% (-0.2%, 0.3%) |
| Opioids; n (%) | 10,208 (30.5%) | 18,282 (31.0%) | -0.5% (-1.1%, 0.2%) | 7,633 (30.8%) | 7,606 (30.7%) | 0.1% (-0.7%, 0.9%) |
| Anti-depressants; n (%) | 13,271 (39.7%) | 23,749 (40.3%) | -0.6% (-1.2%, 0.1%) | 9,848 (39.7%) | 9,931 (40.1%) | -0.3% (-1.2%, 0.5%) |
| Antipsychotics; n (%) | 1,863 (5.6%) | 2,713 (4.6%) | 1.0% (0.7%, 1.3%) | 1,253 (5.1%) | 1,269 (5.1%) | -0.1% (-0.5%, 0.3%) |
| Anxiolytics / hypnotics, benzos; n (%) | 6,681 (20.0%) | 13,427 (22.8%) | -2.8% (-3.3%, -2.2%) | 5,141 (20.7%) | 5,147 (20.8%) | -0.0% (-0.7%, 0.7%) |
| Dementia medications; n (%) | 713 (2.1%) | 632 (1.1%) | 1.1% (0.9%, 1.2%) | 389 (1.6%) | 399 (1.6%) | -0.0% (-0.3%, 0.2%) |
| Urinary tract infections antibiotics; n (%) | 15,139 (45.3%) | 28,224 (47.9%) | -2.6% (-3.2%, -1.9%) | 11,421 (46.1%) | 11,387 (45.9%) | 0.1% (-0.7%, 1.0%) |
| Laxatives: n (%) | 1,259 (3.8%) | 2,046 (3.5%) | 0.3% (0.0%, 0.6%) | 908 (3.7%) | 893 (3.6%) | 0.1% (-0.3%, 0.4%) |
| Number of distinct medications | | | | | | |
| mean (sd) | 15.30 (7.15) | 14.48 (7.21) | 0.82 (0.72, 0.92) | 15.00 (7.15) | 15.03 (7.20) | -0.04 (-0.16, 0.09) |
| median [IQR] | 14.00 [10.00, 19.00] | 13.00 [9.00, 18.00] | - (-, -) | 14.00 [10.00, 19.00] | 14.00 [10.00, 19.00] | - (-, -) |
| min. max | 1.00, 67.00 | 1.00, 69.00 | - (-, -) | 1.00, 67.00 | 1.00, 67.00 | - (-, -) |
| Number of office visits | | , | ,,,, | , | , | ` ' ' |
| mean (sd) | 9.50 (7.07) | 9.67 (7.19) | -0.17 (-0.27, -0.08) | 9.52 (7.15) | 9.55 (6.89) | -0.03 (-0.15, 0.10) |
| median [IQR] | 8.00 [5.00, 13.00] | 8.00 [5.00, 13.00] | - (-, -) | 8.00 [4.00, 13.00] | 8.00 [5.00, 13.00] | - (-, -) |
| min, max | 0.00, 122.00 | 0.00, 94.00 | - (-, -) | 0.00, 122.00 | 0.00, 80.00 | - (-, -) |
| Number of endocrinologist visits | 0.00, 122.00 | 0.00, 54.00 | (, , | 0.00, 122.00 | 0.00, 00.00 | (, , |
| mean (sd) | 0.49 (1.59) | 0.43 (1.41) | 0.07 (0.05, 0.09) | 0.47 (1.50) | 0.48 (1.48) | -0.01 (-0.04, 0.01) |
| median [IOR] | 0.00 [0.00, 0.00] | 0.00 (0.00, 0.00) | - (-, -) | 0.00 (0.00, 0.00) | 0.00 [0.00, 0.00] | - () |
| min, max | 0.00, 53.00 | 0.00, 85.00 | - (-, -) | 0.00, 52.00 | 0.00, 85.00 | - (-, -) |
| Number of cardiologist visits | 0.00, 33.00 | 0.00, 03.00 | ( , ) | 0.00, 32.00 | 0.00, 03.00 | ( , ) |
| mean (sd) | 1.59 (3.61) | 1.49 (3.28) | 0.10 (0.05, 0.15) | 1.51 (3.46) | 1.52 (3.37) | -0.01 (-0.07, 0.05) |
| median [IQR] | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | - (-, -) | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | - (-, -) |
| min, max | 0.00, 97.00 | 0.00, 96.00 | - (-, -) | 0.00, 97.00 | 0.00, 96.00 | - (-, -) |
| Number of internal/family medicine visits | 0.00, 37.00 | 0.00, 30.00 | - (-, -) | 0.00, 37.00 | 0.00, 30.00 | - (-, -) |
| mean (sd) | 7.98 (9.82) | 6.68 (7.50) | 1.30 (1.18, 1.42) | 7.25 (8.38) | 7.28 (8.50) | -0.03 (-0.18, 0.12) |
| median [IQR] | 5.00 [3.00, 9.00] | 5.00 [3.00, 8.00] | - (-, -) | 5.00 [3.00, 9.00] | 5.00 [3.00, 9.00] | - (-, -) |
| min, max | 0.00, 281.00 | 0.00, 225.00 | - (-, -)<br>- (-, -) | 0.00, 156.00 | 0.00, 225.00 | - (-, -)<br>- (-, -) |
| Number of electrocardiograms (ECG/EKG) | 0.00, 281.00 | 0.00, 223.00 | - (-, -) | 0.00, 136.00 | 0.00, 223.00 | - (-, -) |
| mean (sd) | 0.98 (1.73) | 0.90 (1.60) | 0.09 (0.07, 0.11) | 0.92 (1.67) | 0.93 (1.60) | -0.01 (-0.04, 0.02) |
| median [IOR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | - (-, -) | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | - (-, -) |
| min, max | 0.00 [0.00, 1.00] | 0.00, 59.00 | - (-, -)<br>- (-, -) | 0.00, 59.00 | 0.00, 28.00 | - (-, -)<br>- (-, -) |
| Number of echocardiograms | 0.00, 39.00 | 0.00, 39.00 | - (-, -) | 0.00, 39.00 | 0.00, 28.00 | - (-, -) |
| | 0.29 (0.67) | 0.26 (0.60) | 0.03 (0.02, 0.04) | 0.27 (0.66) | 0.27 (0.62) | -0.00 (-0.01, 0.01) |
| mean (sd)median [IQR] | 0.29 (0.07) | 0.00 [0.00, 0.00] | - (-, -) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) |
| min. max | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -)<br>- (-, -) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -)<br>- (-, -) |
| | 0.00, 33.00 | 0.00, 13.00 | - (-, -) | 0.00, 33.00 | 0.00, 10.00 | - (-, -) |
| Out-of-pocket medication cost | COC 2C (0F0 27) | E01 E0 (700 EE) | 24 77 (12 00 25 00) | F00 C0 (072 17) | E00 EE (700 11) | 1.00 / 12.10 15.22 |
| mean (sd) | 606.26 (850.27) | 581.50 (786.55) | 24.77 (13.66, 35.88) | 599.60 (873.17) | 598.55 (729.11) | 1.06 (-13.10, 15.22) |
| median [IQR] | 330.91 [115.80, 821.96] | 330.72 [122.31, 769.78] | - (-, -) | 329.57 [117.42, 805.63] | 346.29 [126.66, 817.82] | - (-, -) |
| min, max | 0.00, 49,246.61 | 0.00, 36,280.29 | - (-, -) | 0.00, 49,246.61 | 0.00, 22,732.61 | - (-, -) |
| Unique brand medicines | | | | | <u> </u> | |
| mean (sd) | 15.60 (7.42) | 14.71 (7.42) | 0.90 (0.80, 1.00) | 15.27 (7.38) | 15.31 (7.44) | -0.03 (-0.17, 0.10) |
| median [IQR] | 14.00 [10.00, 20.00] | 13.00 [9.00, 19.00] | - (-, -) | 14.00 [10.00, 19.00] | 14.00 [10.00, 19.00] | - (-, -) |
| min, max | 1.00, 70.00 | 1.00, 77.00 | - (-, -) | 1.00, 70.00 | 1.00, 70.00 | - (-, -) |
| Unique generic medicines | | | | <u> </u> | <u> </u> | <b>+</b> |
| mean (sd) | 15.30 (7.15) | 14.48 (7.21) | 0.82 (0.72, 0.92) | 15.00 (7.15) | 15.03 (7.20) | -0.04 (-0.16, 0.09) |
| median [IQR] | 14.00 [10.00, 19.00] | 13.00 [9.00, 18.00] | - (-, -) | 14.00 [10.00, 19.00] | 14.00 [10.00, 19.00] | - (-, -) |
| min, max | 1.00, 67.00 | 1.00, 69.00 | - (-, -) | 1.00, 67.00 | 1.00, 67.00 | - (-, -) |
| Colonoscopy Sigmoidoscopy; n (%) | 3,304 (9.9%) | 6,385 (10.8%) | -0.9% (-1.4%, -0.5%) | 2,562 (10.3%) | 2,525 (10.2%) | 0.1% (-0.4%, 0.7%) |
| Flu Pneumococcal vaccine; n (%) | 11,686 (35.0%) | 17,681 (30.0%) | 5.0% (4.3%, 5.6%) | 8,299 (33.5%) | 8,361 (33.7%) | -0.3% (-1.1%, 0.6%) |
| Pap smear, n (%) | 1,813 (5.4%) | 4,598 (7.8%) | -2.4% (-2.7%, -2.0%) | 1,493 (6.0%) | 1,478 (6.0%) | 0.1% (-0.4%, 0.5%) |

| PSA test: n (%) | 6,876 (20.6%) | 13,445 (22.8%) | -2.2% (-2.8%, -1.7%) | 5.317 (21.4%) | 5,378 (21.7%) | -0.2% (-1.0%, 0.5%) |
|---|---|---|---|---|---|---|
| Fecal occult blood test; n (%) | 1,507 (4.5%) | 2,181 (3.7%) | 0.8% (0.5%, 1.1%) | 1,001 (4.0%) | 1,019 (4.1%) | -0.2% (-1.0%, 0.3%) |
| Bone mineral density tests; n (%) | 2,313 (6.9%) | 4,345 (7.4%) | -0.4% (-0.8%, -0.1%) | 1,758 (7.1%) | 1,747 (7.0%) | 0.0% (-0.4%, 0.5%) |
| Mammograms; n (%) | 7,806 (23.4%) | 16,016 (27.2%) | -3.8% (-4.4%, -3.2%) | 6,150 (24.8%) | 6,154 (24.8%) | -0.0% (-0.4%, 0.5%) |
| Telemedicine; n (%) | 7,678 (23.0%) | 14,008 (23.8%) | -0.8% (-1.4%, -0.2%) | 5,591 (22.5%) | 5,648 (22.8%) | -0.2% (-1.0%, 0.5%) |
| HbA1c tests | 7,678 (23.0%) | 14,008 (23.8%) | -0.8% (-1.4%, -0.2%) | 5,591 (22.5%) | 5,646 (22.6%) | -0.2% (-1.0%, 0.5%) |
| | 0.47.(4.00) | 0.00 (4.04) | 0.10 (0.10, 0.00) | 0.44./4.00 | 0.40.(1.20) | 0.01 / 0.02 0.00 |
| mean (sd) | 2.47 (1.38) | 2.29 (1.31) | 0.18 (0.16, 0.20) | 2.41 (1.32) | 2.42 (1.39) | -0.01 (-0.03, 0.02) |
| median [IQR] | 2.00 [2.00, 3.00] | 2.00 [1.00, 3.00] | - (-, -) | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | - (-, -) |
| min, max | 0.00, 40.00 | 0.00, 44.00 | - (-, -) | 0.00, 26.00 | 0.00, 44.00 | - (-, -) |
| Lipid panels | | | | | | |
| mean (sd) | 1.57 (1.15) | 1.64 (1.14) | -0.07 (-0.09, -0.06) | 1.59 (1.15) | 1.61 (1.14) | -0.01 (-0.03, 0.01) |
| median [IQR] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | - (-, -) | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | - (-, -) |
| min, max | 0.00, 26.00 | 0.00, 26.00 | - (-, -) | 0.00, 26.00 | 0.00, 26.00 | - (-, -) |
| Creatinine tests | | | | | | |
| mean (sd) | 3.08 (3.07) | 2.76 (2.80) | 0.32 (0.28, 0.36) | 2.93 (2.74) | 2.95 (3.07) | -0.02 (-0.07, 0.03) |
| median [IQR] | 2.00 [1.00, 4.00] | 2.00 [1.00, 4.00] | - (-, -) | 2.00 [1.00, 4.00] | 2.00 [1.00, 4.00] | - (-, -) |
| min, max | 0.00, 85.00 | 0.00, 105.00 | - (-, -) | 0.00, 73.00 | 0.00, 105.00 | - (-, -) |
| Natriuretic peptide tests | | | | | | |
| mean (sd) | 0.20 (0.83) | 0.17 (0.69) | 0.03 (0.02, 0.04) | 0.18 (0.70) | 0.18 (0.72) | -0.00 (-0.02, 0.01) |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) |
| min, max | 0.00, 68.00 | 0.00, 28.00 | - (-, -) | 0.00, 28.00 | 0.00, 27.00 | - (-, -) |
| Urine tests | | | | | | |
| mean (sd) | 1.05 (1.66) | 1.03 (1.62) | 0.02 (-0.00, 0.04) | 1.03 (1.66) | 1.03 (1.60) | -0.00 (-0.03, 0.03) |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | - (-, -) | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | - (-, -) |
| min, max | 0.00, 34.00 | 0.00, 37.00 | - (-, -) | 0.00, 34.00 | 0.00, 37.00 | - (-, -) |
| Combined comorbidity score | | | | | | |
| mean (sd) | 2.30 (2.60) | 1.80 (2.28) | 0.50 (0.47, 0.53) | 2.06 (2.40) | 2.08 (2.45) | -0.02 (-0.06, 0.02) |
| median [IQR] | 2.00 [0.00, 4.00] | 1.00 [0.00, 3.00] | - (-, -) | 1.00 [0.00, 3.00] | 1.00 [0.00, 3.00] | - (-, -) |
| min, max | -2.00, 16.00 | -2.00, 16.00 | - (-, -) | -2.00, 16.00 | -2.00, 16.00 | - (-, -) |
| Frailty Score | | | | | Ì | |
| mean (sd) | 0.17 (0.06) | 0.16 (0.05) | 0.01 (0.01, 0.01) | 0.17 (0.06) | 0.17 (0.06) | -0.00 (-0.00, 0.00) |
| median [IQR] | 0.16 [0.13, 0.20] | 0.15 [0.13, 0.19] | - (-, -) | 0.16 [0.13, 0.20] | 0.16 [0.13, 0.20] | - (-, -) |
| min, max | 0.05, 0.57 | 0.04, 0.62 | - (-, -) | 0.06, 0.57 | 0.04, 0.62 | - (-, -) |
| Number of Hospitalizations | 0.00, 0.07 | 0.0 1, 0.02 | (, ) | 0.00, 0.07 | 5.5 1, 5.52 | |
| mean (sd) | 0.27 (0.84) | 0.16 (0.58) | 0.10 (0.09, 0.11) | 0.21 (0.68) | 0.21 (0.69) | -0.00 (-0.01, 0.01) |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) |
| min, max | 0.00, 20.00 | 0.00, 12.00 | - (-, -) | 0.00, 17.00 | 0.00, 12.00 | - (-, -) |
| Any hospitalization within prior 91 days; n (%) | 1,980 (5.9%) | 2,078 (3.5%) | 2.4% (2.1%, 2.7%) | 1,115 (4.5%) | 1,150 (4.6%) | -0.1% (-0.5%, 0.2%) |
| Any hospitalization within prior 92-365 days; n (%) | 3,936 (11.8%) | 5,169 (8.8%) | 3.0% (2.6%, 3.4%) | 2,519 (10.2%) | 2,480 (10.0%) | 0.2% (-0.4%, 0.7%) |
| Number of hospitalizations (0, 1, 2 or more) | 3,930 (11.670) | 3,103 (6.670) | 3.0% (2.6%, 3.4%) | 2,519 (10.270) | 2,480 (10.0%) | 0.270 (-0.470, 0.770) |
| <1; n (%) | 28,313 (84.7%) | 52,488 (89.0%) | -4.3% (-4.8%, -3.8%) | 21,595 (87.1%) | 21,608 (87.1%) | -0.1% (-0.6%, 0.5%) |
| | | · · · · · · | | | | |
| 1 - <2; n (%) | 3,216 (9.6%) | 4,588 (7.8%) | 1.8% (1.5%, 2.2%) | 2,165 (8.7%) | 2,150 (8.7%) | 0.1% (-0.4%, 0.6%) |
| >= 2; n (%) | 1,891 (5.7%) | 1,879 (3.2%) | 2.5% (2.2%, 2.8%) | 1,035 (4.2%) | 1,037 (4.2%) | -0.0% (-0.4%, 0.3%) |
| Heart failure hospitalization; n (%) | 1,492 (4.5%) | 1,714 (2.9%) | 1.6% (1.3%, 1.8%) | 904 (3.6%) | 901 (3.6%) | 0.0% (-0.3%, 0.3%) |
| ED visit; n (%) | 10,963 (32.8%) | 15,564 (26.4%) | 6.4% (5.8%, 7.0%) | 7,464 (30.1%) | 7,453 (30.1%) | 0.0% (-0.8%, 0.9%) |
| Acute MI; n (%) | 430 (1.3%) | 482 (0.8%) | 0.5% (0.3%, 0.6%) | 268 (1.1%) | 264 (1.1%) | 0.0% (-0.2%, 0.2%) |
| Old MI; n (%) | 1,769 (5.3%) | 2,189 (3.7%) | 1.6% (1.3%, 1.9%) | 1,143 (4.6%) | 1,142 (4.6%) | 0.0% (-0.4%, 0.4%) |
| Heart failure; n (%) | 5,287 (15.8%) | 7,343 (12.5%) | 3.4% (2.9%, 3.8%) | 3,514 (14.2%) | 3,572 (14.4%) | -0.2% (-0.9%, 0.4%) |
| Acute heart failure; n (%) | 1,374 (4.1%) | 1,674 (2.8%) | 1.3% (1.0%, 1.5%) | 861 (3.5%) | 872 (3.5%) | -0.0% (-0.4%, 0.3%) |
| Microalbuminuria or proteinuria; n (%) | 2,630 (7.9%) | 3,606 (6.1%) | 1.8% (1.4%, 2.1%) | 1,813 (7.3%) | 1,811 (7.3%) | 0.0% (-0.5%, 0.5%) |
| Ratio of brand to generic medications | | | | | | |
| mean (sd) | 1.02 (0.04) | 1.01 (0.04) | 0.00 (0.00, 0.00) | 1.02 (0.04) | 1.02 (0.04) | -0.00 (-0.00, 0.00) |
| median [IQR] | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | - (-, -) | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | - (-, -) |
| min, max | 0.79, 1.50 | 0.80, 1.50 | - (-, -) | 0.90, 1.50 | 0.88, 1.50 | - (-, -) |

| MARKETSCAN<br>Variable | Reference: Dulaglutide | Exposure: Tirzepatide | Difference | Reference: Dulaglutide | Exposure: Tirzepatide | Difference |
|---|---|---|---|---|---|---|
| Number of patients<br>Year of Cohort Entry Date | 19,927 | 23,787 | 17.7 | 14,357 | 14,357 | - (-, -) |
| _2022; n(%) | 8,893 (44.6%) | 4,332 (18.2%) | 26.4% (25.6%, 27.3%) | 4,180 (29.1%) | 4,181 (29.1%) | -0.0% (-11%,11%) |
| _2023; n(%) | 11,034 (55.4%) | 19,455 (81.8%) | -26.4% (-27.3%, -25.6% | 10,177 (70.9%) | 10,176 (70.9%) | 0.0% (-11%,11%) |
| Age _mean (sd) | 56.41 (11.05) | 53.84 (10.02) | 2.58 (2.38, 2.78) | 55.00 (10.54) | 55.04 (10.15) | -0.03 (-0.27, 0.21) |
| _median [IQR] _min_max | 57.00 [49.00,63.00]<br>18.00,95.00 | 54.00 [48.00,60.00]<br>18.00,96.00 | - (-, -)<br>- (-, -) | 55.00 [48.00, 62.00]<br>18.00, 91.00<br>6.711 (46.7%) | 55.00 [49.00, 61.00]<br>19.00, 96.00 | - (-, -)<br>- (-, -) |
| Gender (male); n (%)<br>Region / State<br>Northeast; n (%) | 9,695 (48.7%)<br>2,386 (12.0%) | 10,568 (44.4%) | 4.2% (3.3%, 5.2%)<br>3.3% (2.7%, 3.9%) | 1,485 (10.3%) | 6,745 (47.0%)<br>1,499 (10.4%) | -0.2% (-1.4%, 0.9%)<br>-0.1% (-0.8%, 0.6%) |
| _Widwest / North central; n (%) | 6,172 (31.0%) | 5,247 (22.1%) | 8.9% (8.1%, 9.7%) | 3,881 (27.0%) | 3,807 (26.5%) | 0.5% (-0.5%, 1.5%) |
| _South: n (%) | 9,614 (48.2%) | 14,692 (61.8%) | -13.5% (-14.5%, -12.6%) | | 7.838 (54.6%) | -0.5% (-1.7%, 0.6%) |
| | 1,740 (8.7%) | 1,765 (7.4%) | 1.3% (0.8%, 1.8%) | 1,222 (8.5%) | 1,201 (8.4%) | 0.1% (-0.5%, 0.8%) |
| | 15 (0.1%) | 18 (0.1%) | -0.0% (-0.1%, 0.1%) | 9 (0.1%) | 12 (0.1%) | -0.0% (-0.1%, 0.0%) |
| Smoking / Tobacco use; n (%) Weight | 2,192 (11.0%) | 2,227 (9.4%) | 1.6% (1.1%, 2.2%) | 1,462 (10.2%) | 1,459 (10.2%) | 0.0% (-0.7%, 0.7%) |
| _Overweight; n (%) | 2,417 (12.1%) | 1,845 (7.8%) | 4.4% (3.8%, 4.9%) | 1,388 (9.7%) | 1,393 (9.7%) | -0.0% (-0.7%, 0.7%) |
| _Class 1 Obesity; n (%) | 1,925 (9.7%) | 1,862 (7.8%) | 1.8% (1.3%, 2.4%) | 1,237 (8.6%) | 1,235 (8.6%) | 0.0% (-0.6%, 0.7%) |
| _Class 2 Obesity; n (%) | 1,322 (6.6%) | 1,634 (6.9%) | -0.2% (-0.7%, 0.2%) | 991 (6.9%) | 1,003 (7.0%) | -0.1% (-0.7%, 0.5%) |
| _Class 3 Obesity; n (%) | 5,184 (26.0%) | 5,167 (21.7%) | 4.3% (3.5%, 5.1%) | 3,453 (24.1%) | 3,414 (23.8%) | 0.3% (-0.7%, 1.3%) |
| _Unspecified Obesity; n (%) Diabetic retinopathy; n (%) | 9,079 (45.6%) | 13,279 (55.8%) | -10.3% (-11.2%, -9.3%) | 7,288 (50.8%) | 7,312 (50.9%) | -0.2% (-1.3%,1.0%) |
| | 1,551 (7.8%) | 1,229 (5.2%) | 2.6% (2.1%, 3.1%) | 929 (6.5%) | 934 (6.5%) | -0.0% (-0.6%, 0.5%) |
| Diabetic neuropathy; n (%) Diabetic nephropathy; n (%) | 3,742 (18.8%) | 3,133 (13.2%) | 5.6% (4.9%, 6.3%) | 2,248 (15.7%) | 2,316 (16.1%) | -0.5% (-1.3%, 0.4%) |
| | 2,932 (14.7%) | 2,385 (10.0%) | 4.7% (4.1%, 5.3%) | 1,711 (11.9%) | 1,754 (12.2%) | -0.3% (-1.1%, 0.5%) |
| Diabetes with other opthalmic complications; n (%) Diabetes with peripheral circulatory disorders; n (%) | 331 (1.7%)<br>1,726 (8.7%) | 294 (1.2%)<br>1,643 (6.9%)<br>313 (1.3%) | 0.4% (0.2%, 0.7%)<br>1.8% (1.2%, 2.3%)<br>0.7% (0.4%, 0.9%) | 214 (1.5%)<br>1,072 (7.5%)<br>226 (1.6%) | 221 (1.5%)<br>1,120 (7.8%)<br>231 (1.6%) | -0.0% (-0.3%, 0.2%)<br>-0.3% (-1.0%, 0.3%)<br>-0.0% (-0.3%, 0.3%) |
| Diabetic foot; n (%) Erectile dysfunction; n (%) Hypoglycemia; n (%) | 394 (2.0%)<br>742 (3.7%)<br>3,641 (18.3%) | 798 (3.4%)<br>4.310 (18.1%) | 0.4% (0.0%, 0.7%) | 539 (3.8%)<br>2,587 (18.0%) | 540 (3.8%)<br>2,623 (18.3%) | -0.0% (-0.5%, 0.4%)<br>-0.3% (-11%, 0.6%) |
| Hyperglycemia, II(%) Hyperglycemia/DKA/HONK; n(%) Skininfections; n(%) | 10,889 (54.6%) | 11,497 (48.3%) | 6.3% (5.4%, 7.3%) | 7,460 (52.0%) | 7,496 (52.2%) | -0.3% (-1.4%, 0.9%) |
| | 1,889 (9.5%) | 2,027 (8.5%) | 1.0% (0.4%, 1.5%) | 1,264 (8.8%) | 1,312 (9.1%) | -0.3% (-1.0%, 0.3%) |
| Stable angina; n (%) Unstable angina; n (%) | 506 (2.5%) | 425 (1.8%) | 0.8% (0.5%, 1.0%) | 291 (2.0%) | 306 (2.1%) | -0.1% (-0.4%, 0.2%) |
| | 343 (1.7%) | 271 (1.1%) | 0.6% (0.4%, 0.8%) | 193 (1.3%) | 197 (1.4%) | -0.0% (-0.3%, 0.2%) |
| Hypertension; n (%) | 16,057 (80.6%) | 19,082 (80.2%) | 0.4% (-0.4%,1.1%) | 11,463 (79.8%) | 11,494 (80.1%) | -0.2% (-1.1%, 0.7%) |
| Hypotension; n (%) | 315 (1.6%) | 252 (1.1%) | 0.5% (0.3%, 0.7%) | 165 (1.1%) | 170 (1.2%) | -0.0% (-0.3%, 0.2%) |
| Hyperlipidemia; n (%) | 15,727 (78.9%) | 18,587 (78.1%) | 0.8% (0.0%, 1.6%) | 11,299 (78.7%) | 11,319 (78.8%) | -0.1% (-1.1%, 0.8%) |
| Atrial fibrillation; n (%) | 1,181 (5.9%) | 1,059 (4.5%) | 1.5% (1.1%, 1.9%) | 724 (5.0%) | 724 (5.0%) | 0.0% (-0.5%, 0.5%) |
| Cardiac conduction disorder; n (%) Previous cardiac procedure (CABG, PTCA, Stent); n (%) | 678 (3.4%) | 572 (2.4%) | 1.0% (0.7%, 1.3%) | 388 (2.7%) | 401 (2.8%) | -0.1% (-0.5%, 0.3%) |
| | 268 (1.3%) | 210 (0.9%) | 0.5% (0.3%, 0.7%) | 159 (1.1%) | 152 (1.1%) | 0.0% (-0.2%, 0.3%) |
| Ischemic stroke; n (%) PVD diagnosis or surgery; n (%) | 200 (1.0%) | 124 (0.5%) | 0.5% (0.3%, 0.7%) | 97 (0.7%) | 104 (0.7%) | -0.0% (-0.2%, 0.2%) |
| | 916 (4.6%) | 781 (3.3%) | 1.3% (0.9%, 1.7%) | 526 (3.7%) | 550 (3.8%) | -0.2% (-0.6%, 0.3%) |
| Other cardiac dysrhythmia; n (%) Cardiomyopathy; n (%) | 2,854 (14.3%) | 3,151 (13.2%) | 1.1% (0.4%, 1.7%) | 1,889 (13.2%) | 1,925 (13.4%) | -0.3% (-1.0%, 0.5%) |
| | 628 (3.2%) | 571 (2.4%) | 0.8% (0.4%, 1.1%) | 379 (2.6%) | 379 (2.6%) | 0.0% (-0.4%, 0.4%) |
| Valve disorders; n (%) Valve replacement; n (%) | 1,242 (6.2%) | 1,229 (5.2%) | 1.1% (0.6%, 1.5%) | 793 (5.5%) | 814 (5.7%) | -0.1% (-0.7%, 0.4%) |
| | 113 (0.6%) | 82 (0.3%) | 0.2% (0.1%, 0.4%) | 61 (0.4%) | 60 (0.4%) | 0.0% (-0.1%, 0.2%) |
| TIA; n (%)<br>Edema; n (%) | 232 (1.2%)<br>1,531 (7.7%) | 211 (0.9%)<br>1,669 (7.0%) | 0.3% (0.1%, 0.5%)<br>0.7% (0.2%, 1.2%)<br>0.4% (0.1%, 0.7%) | 137 (1.0%)<br>983 (6.8%) | 140 (1.0%)<br>1,020 (7.1%) | -0.0% (-0.3%, 0.2%)<br>-0.3% (-0.9%, 0.3%) |
| Venous thromboembolism / Pulmonary embolism; n (%) Pulmonary hypertension; n (%) Implantable cardioverter defibrillator; n (%) | 488 (2.4%)<br>232 (1.2%)<br>45 (0.2%) | 483 (2.0%)<br>226 (1.0%)<br>32 (0.1%) | 0.2% (0.0%, 0.4%) | 322 (2.2%)<br>149 (1.0%)<br>20 (0.1%) | 327 (2.3%)<br>143 (1.0%)<br>24 (0.2%) | -0.0% (-0.4%, 0.3%)<br>0.0% (-0.2%, 0.3%)<br>-0.0% (-0.1%, 0.1%) |
| Hyperkalemia; n (%) Coronary atherosclerosis: n (%) | 330 (1.7%)<br>2.522 (12.7%) | 236 (1.0%)<br>2.320 (9.8%) | 0.7% (0.4%, 0.9%) | 158 (1.1%)<br>1.552 (10.8%) | 178 (1.2%)<br>1.592 (11.1%) | -0.0% (-0.1%, 0.1%)<br>-0.1% (-0.4%, 0.1%)<br>-0.3% (-1.0%, 0.5%) |
| Cerebrovascular procedure; n (%) Insertion of pacemakers / removal of cardiac lead; n (%) | 14 (0.1%)<br>15 (0.1%) | 9 (0.0%)<br>7 (0.0%) | 0.0% (-0.0%, 0.1%) | 6 (0.0%)<br>7 (0.0%) | 8 (0.1%)<br>6 (0.0%) | -0.0% (-0.1%, 0.0%)<br>0.0% (-0.0%, 0.1%) |
| CKD stage 1-2; n (%) | 411 (2.1%) | 485 (2.0%) | 0.0% (-0.2%, 0.3%) | 288 (2.0%) | 292 (2.0%) | -0.0% (-0.4%, 0.3%) |
| CKD stage 3-4; n (%) | 1,440 (7.2%) | 1,006 (4.2%) | 3.0% (2.6%, 3.4%) | 738 (5.1%) | 764 (5.3%) | -0.2% (-0.7%, 0.3%) |
| Unspecified CKD; n (%) | 465 (2.3%) | 352 (1.5%) | 0.9% (0.6%, 1.1%) | 249 (1.7%) | 263 (1.8%) | -0.1% (-0.4%, 0.2%) |
| Acute kidney injury; n (%) | 781 (3.9%) | 575 (2.4%) | 1.5% (1.2%, 1.8%) | 395 (2.8%) | 420 (2.9%) | -0.2% (-0.6%, 0.2%) |
| Hypertensive nephropathy; n (%) Urinary tract infections; n (%) | 1,215 (6.1%) | 984 (4.1%) | 2.0% (1.5%, 2.4%) | 678 (4.7%) | 701 (4.9%) | -0.2% (-0.7%, 0.3%) |
| | 1,775 (8.9%) | 2,209 (9.3%) | -0.4% (-0.9%, 0.2%) | 1,254 (8.7%) | 1,228 (8.6%) | 0.2% (-0.5%, 0.8%) |
| Genital infections; n (%) | 818 (4.1%) | 868 (3.6%) | 0.5% (0.1%, 0.8%) | 560 (3.9%) | 570 (4.0%) | -0.1% (-0.5%, 0.4%) |
| Urolithiasis (Kidney and urinary stone); n (%) | 802 (4.0%) | 934 (3.9%) | 0.1% (-0.3%, 0.5%) | 568 (4.0%) | 557 (3.9%) | 0.1% (-0.4%, 0.5%) |
| COPD; n (%) | 993 (5.0%) | 885 (3.7%) | 1.3% (0.9%, 1.7%) | 578 (4.0%) | 1,291 (9.0%) | -0.2% (-0.7%, 0.3%) |
| Asthma; n (%) | 1,730 (8.7%) | 2,194 (9.2%) | -0.5% (-1.1%, -0.0%) | 1,262 (8.8%) | | -0.2% (-0.9%, 0.5%) |
| Obstructive sleep apnea; n (%) Serious bacterial infections; n (%) | 5,350 (26.8%) | 7,089 (29.8%) | -3.0% (-3.8%, -2.1%) | 3,983 (27.7%) | 4,021 (28.0%) | -0.3% (-1.3%, 0.8%) |
| | 617 (3.1%) | 505 (2.1%) | 1.0% (0.7%, 1.3%) | 354 (2.5%) | 370 (2.6%) | -0.1% (-0.5%, 0.3%) |
| Pneumonia; n(%) | 683 (3.4%) | 626 (2.6%) | 0.8% (0.5%, 11%) | 398 (2.8%) | 411 (2.9%) | -0.1% (-0.5%, 0.3%) |
| Liver disease; n (%) | 2,583 (13.0%) | 3,297 (13.9%) | -0.9% (-1.5%, -0.3%) | 1,875 (13.1%) | 1,883 (13.1%) | -0.1% (-0.8%, 0.7%) |
| MASH/MASLD; n (%) | 1,583 (7.9%) | 2,216 (9.3%) | -1.4% (-1.9%, -0.8%) | 1,212 (8.4%) | 1,219 (8.5%) | -0.0% (-0.7%, 0.6%) |
| MASH/MASLU; II (%) Fractures / Falls; n (%) Osteoporosis; n (%) | 743 (3.7%)<br>273 (1.4%) | 2,216 (9.5%)<br>687 (2.9%)<br>273 (1.1%) | 0.8% (0.5%, 1.2%) | 459 (3.2%)<br>186 (1.3%) | 461 (3.2%)<br>180 (1.3%) | -0.0% (-0.4%, 0.4%)<br>-0.0% (-0.2%, 0.3%) |
| Osteoarthritis; n (%) Depression; n (%) | 3,860 (19.4%)<br>3.114 (15.6%) | 4,531 (19.0%)<br>3,706 (15.6%) | 0.3% (-0.4%,11%) | 2,725 (19.0%)<br>2,226 (15.5%) | 2,719 (18.9%)<br>2,236 (15.6%) | 0.0% (-0.9%, 1.0%) |
| Dementia; n (%) Delirium or psychosis; n (%) | 311 (1.6%)<br>140 (0.7%) | 147 (0.6%)<br>85 (0.4%) | 0.9% (0.7%, 1.1%) | 116 (0.8%)<br>67 (0.5%) | 119 (0.8%)<br>73 (0.5%) | -0.0% (-0.2%, 0.2%)<br>-0.0% (-0.2%, 0.1%) |
| Anxiety; n (%) | 3,610 (181%) | 4,986 (21.0%) | -2.8% (-3.6%, -2.1%) | 2,708 (18.9%) | 2,770 (19.3%) | -0.4% (-1.3%, 0.5%) |
| Sleep disorders; n (%) | 4,422 (22.2%) | 5,954 (25.0%) | -2.8% (-3.6%, -2.0%) | 3,346 (23.3%) | 3,328 (23.2%) | 0.1% (-0.9%, 1.1%) |
| Anemia; n (%) | 2,717 (13.6%) | 3,294 (13.8%) | -0.2% (-0.9%, 0.4%) | 1,872 (13.0%) | 1,931 (13.4%) | -0.4% (-1.2%, 0.4%) |
| Influenza; n (%) | 295 (1.5%) | 602 (2.5%) | -1.1% (-1.3%, -0.8%) | 254 (1.8%) | 272 (1.9%) | -0.1% (-0.4%, 0.2%) |
| COVID; n(%) Hyperthyroidism and other thyroid gland disorders; n(%) | 2,752 (13.8%)<br>3,904 (19.6%) | 3,133 (13.2%)<br>5,303 (22.3%) | 0.6% (-0.0%, 1.3%)<br>-2.7% (-3.5%, -1.9%) | 1,920 (13.4%)<br>2,881 (20.1%) | 1,893 (13.2%)<br>2,902 (20.2%) | 0.2% (-0.6%, 1.0%) -0.1% (-1.1%, 0.8%) |
| Hypothyroidism; n (%) Nephrotic syndrome; n (%) | 3,023 (15.2%) | 4,153 (17.5%) | -2.3% (-3.0%, -1.6%) | 2,246 (15.6%) | 2,282 (15.9%) | -0.3% (-11%, 0.6%) |
| | 15 (0.1%) | 8 (0.0%) | 0.0% (-0.0%, 0.1%) | 6 (0.0%) | 7 (0.0%) | -0.0% (-0.1%, 0.0%) |
| Urinary incontinence; n (%) Biliary disease; n (%) | 539 (2.7%)<br>63 (0.3%) | 605 (2.5%)<br>57 (0.2%) | 0.2% (-0.1%, 0.5%) 0.1% (-0.0%, 0.2%) | 373 (2.6%)<br>34 (0.2%) | 388 (2.7%)<br>38 (0.3%) | -0.1% (-0.5%, 0.3%)<br>-0.0% (-0.2%, 0.1%) |
| Pancreatitis; n (%) Bowel obstruction; n (%) Contractorism (%) | 27 (0.1%) | 28 (0.1%) | 0.0% (-0.1%, 0.1%) | 14 (0.1%) | 18 (0.1%) | -0.0% (-0.1%, 0.1%) |
| | 28 (0.1%) | 31 (0.1%) | 0.0% (-0.1%, 0.1%) | 19 (0.1%) | 21 (0.1%) | -0.0% (-0.1%, 0.1%) |
| | 116 (0.6%) | 128 (0.5%) | 0.0% (-0.1%, 0.2%) | 81 (0.6%) | 76 (0.5%) | 0.0% (-0.1%, 0.2%) |
| Gastroparesis; n (%) Number of antidiabetic drugs on CEDmean (sd) | 2.26(1.01) | 2.05 (0.98) | 0.20 (0.18, 0.22) | 2.18 (0.98) | 2.18 (1.02) | 0.00 (-0.02, 0.03) |
| _median[IQR] | 2.00 [2.00, 3.00] | 2.00 [1.00, 3.00] | - (-, -) | 2.00 [1.00, 3.00] | 2.00 [1.00, 3.00] | - (-, -) |
| _min_max | 1.00.6.00 | 1.00, 7.00 | - (-, -) | 1.00, 6.00 | 1.00, 7.00 | - (-, -) |
| Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) | 10,664 (53.5%)<br>3.820 (19.2%) | 11,961 (50.3%)<br>3,213 (13.5%) | 3.2% (2.3%, 4.2%)<br>5.7% (5.0%, 6.4%) | 7,618 (53.1%)<br>2,364 (16.5%) | 7,603 (53.0%)<br>2,388 (16.6%) | 0.1% (-1.1%, 1.3%) |
| Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of DPP-4i; n (%) | 3,509 (17.6%) | 2,591 (10.9%) | 6.7% (6.1%, 7.4%) | 2,057 (14.3%) | 2,043 (14.2%) | 0.1% (-0.7%, 0.9%) |
| | 1,667 (8.4%) | 1,558 (6.5%) | 1.8% (1.3%, 2.3%) | 1,088 (7.6%) | 1,083 (7.5%) | 0.0% (-0.6%, 0.7%) |
| Concomitant use or initiation of SGLT-2i; n(%) Concomitant use or initiation of Any other glucose-lowering drugs; n | 4,397 (22.1%)<br>953 (4.8%) | 4,799 (20.2%)<br>925 (3.9%) | 1.9% (1.1%, 2.7%)<br>0.9% (0.5%, 1.3%) | 3,184 (22.2%)<br>647 (4.5%) | 3,143 (21.9%)<br>656 (4.6%) | 0.3% (-0.7%,1.3%) -0.1% (-0.6%,0.4%) |
| Pastuse of Metformin; n (%) Pastuse of Insulins; n (%) | 14,310 (71.8%) | 16,220 (68.2%) | 3.6% (2.8%, 4.5%) | 10,181 (70.9%) | 10,176 (70.9%) | 0.0% (-1.0%, 1.1%) |
| | 5,321 (26.7%) | 4,504 (18.9%) | 7.8% (7.0%, 8.6%) | 3,264 (22.7%) | 3,317 (23.1%) | -0.4% (-1.3%, 0.6%) |
| Pastuse of Sulfonylureas; n (%) Pastuse of DPP-4l; n (%) | 5,000 (25.1%) | 3,870 (16.3%) | 8.8% (8.1%, 9.6%) | 2,975 (20.7%) | 2,989 (20.8%) | -0.1% (-1.0%, 0.8%) |
| | 2,711 (13.6%) | 2,489 (10.5%) | 3.1% (2.5%, 3.8%) | 1,751 (12.2%) | 1,746 (12.2%) | 0.0% (-0.7%, 0.8%) |
| Pastuse of SGLT-2i; n (%) Pastuse of Any other glucose-lowering drugs; n (%) | 5,884 (29.5%)<br>1,402 (7.0%) | 6,315 (26.5%)<br>1,334 (5.6%) | 3.0% (2.1%, 3.8%)<br>1.4% (1.0%, 1.9%) | 4,175 (29.1%)<br>921 (6.4%) | 4,140 (28.8%)<br>938 (6.5%) | 0.2% (-0.8%,1.3%) -0.1% (-0.7%,0.5%) |
| ACE-is/ARB's; n (%) | 14,316 (71.8%) | 16,441 (69.1%) | 2.7% (1.9%, 3.6%) | 10,121 (70.5%) | 10,123 (70.5%) | -0.0% (-1.1%, 1.0%) |
| ARNI; n (%) | 260 (1.3%) | 272 (1.1%) | 0.2% (-0.1%, 0.4%) | 179 (1.2%) | 169 (1.2%) | 0.1% (-0.2%, 0.3%) |
| Thiazides: n (%) | 6,587 (33.1%) | 8,364 (35.2%) | -2.1% (-3.0%, -1.2%) | 4,843 (33.7%) | 4,832 (33.7%) | 0.1% (-1.0%, 1.2%) |
| Iniazides; n (%) Beta-blockers; n (%) Calcium channel blockers: n (%) | 6,831 (34.3%)<br>5,750 (28.9%) | 7,500 (31.5%)<br>6,445 (27.1%) | 2.8% (1.9%, 3.6%)<br>1.8% (0.9%, 2.6%) | 4,843 (33.7%)<br>4,592 (32.0%)<br>3,976 (27.7%) | 4,832 (33.7%)<br>4,644 (32.3%)<br>3,993 (27.8%) | -0.4% (-1.4%, 0.7%)<br>-0.1% (-1.2%, 0.9%) |
| Calcium chamiei blockers; n(%) Digoxin / Digitoxin, n(%) Loop diuretics; n(%) | 83 (0.4%) | 70 (0.3%) | 0.1% (0.0%, 0.2%) | 49 (0.3%) | 44 (0.3%) | 0.0% (-0.1%, 0.2%) |
| | 2,134 (10.7%) | 2.169 (9.1%) | 1.6% (1.0%, 2.2%) | 1,312 (9.1%) | 1.404 (9.8%) | -0.6% (-1.3%, 0.0%) |
| Other diuretics; n (%) Intravenous diuretics; n (%) | 1,505 (7.6%)<br>153 (0.8%) | 1,773 (7.5%)<br>113 (0.5%) | 0.1% (-0.4%, 0.6%) | 1,073 (7.5%)<br>81 (0.6%) | 1,059 (7.4%)<br>82 (0.6%) | 0.1% (-0.5%, 0.7%)<br>-0.0% (-0.2%, 0.2%) |
| Nitrates; n (%) Anti-arrhythmics; n (%) | 893 (4.5%) | 727 (3.1%) | 1.4% (1.1%, 1.8%) | 522 (3.6%) | 527 (3.7%) | -0.0% (-0.5%, 0.4%) |
| | 284 (1.4%) | 311 (1.3%) | 0.1% (-0.1%, 0.3%) | 197 (1.4%) | 177 (1.2%) | -0.1% (-0.1%, 0.4%) |
| Statins; n (%) PCSK9 inhibitors and other lipid-lowering drugs; n (%) | 15,366 (77.1%) | 16,717 (70.3%) | 6.8% (6.0%, 7.7%) | 10,698 (74.5%) | 10,702 (74.5%) | -0.0% (-1.0%, 1.0%) |
| | 2,478 (12.4%) | 2,820 (11.9%) | 0.6% (-0.0%, 1.2%) | 1,764 (12.3%) | 1,781 (12.4%) | -0.1% (-0.9%, 0.6%) |
| Antiplatelet medications; n (%) Oral anticoagulants; n (%) | 1,882 (9.4%) | 1,673 (7.0%) | 2.4% (1.9%, 2.9%) | 1,169 (8.1%) | 1,161 (8.1%) | 0.1% (-0.6%, 0.7%) |
| | 1,472 (7.4%) | 1,390 (5.8%) | 1.5% (1.1%, 2.0%) | 924 (6.4%) | 921 (6.4%) | 0.0% (-0.6%, 0.6%) |
| COPD/Asthma medications; n (%) | 6,107 (30.6%) | 7,946 (33.4%) | -2.8% (-3.6%, -1.9%) | 4,513 (31.4%) | 4,586 (31.9%) | -0.5% (-1.6%, 0.6%) |
| NSAIDS; n(%) | 6,295 (31.6%) | 8,330 (35.0%) | -3.4% (-4.3%, -2.5%) | 4,731 (33.0%) | 4,750 (33.1%) | -0.1% (-1.2%, 1.0%) |
| Oral corticosteroids; n (%) Osteoporosis agents (incl. bisphosphonates); n (%) | 4,754 (23.9%)<br>309 (1.6%) | 6,781 (28.5%)<br>299 (1.3%) | -4.7% (-5.5%, -3.8%)<br>0.3% (0.1%, 0.5%) | 3,637 (25.3%)<br>202 (1.4%) | 3,629 (25.3%)<br>208 (1.4%) | 0.1% (-1.0%, 1.1%) -0.0% (-0.3%, 0.2%) |
| Opioids; n (%) Anti-depressants; n (%) | 4,830 (24.2%) | 6,002 (25.2%) | -1.0% (-1.8%, -0.2%) | 3,494 (24.3%) | 3,516 (24.5%) | -0.2% (-1.2%, 0.8%) |
| | 6,782 (34.0%) | 8,781 (36.9%) | -2.9% (-3.8%, -2.0%) | 5,030 (35.0%) | 5,111 (35.6%) | -0.6% (-1.7%, 0.5%) |
| Antipsychotics; n(%) Anxiolytics / hypnotics, benzos; n(%) | 576 (2.9%) | 702 (3.0%) | -0.1% (-0.4%, 0.3%) | 407 (2.8%) | 419 (2.9%) | -0.1% (-0.5%, 0.3%) |
| | 3,477 (17.4%) | 5,012 (21.1%) | -3.6% (-4.4%, -2.9%) | 2,679 (18.7%) | 2,723 (19.0%) | -0.3% (-1.2%, 0.6%) |

| Dementia medications; n (%) | 153 (0.8%) | 55 (0.2%) | 0.5% (0.4%, 0.7%) | 44 (0.3%) | 49 (0.3%) | -0.0% (-0.2%, 0.1%) |
|---|---|---|---|---|---|---|
| Urinary tract infections antibiotics: n (%) | 8,510 (42.7%) | 11.083 (46.6%) | -3.9% (-4.8%, -2.9%) | 6,332 (44.1%) | 6,299 (43.9%) | 0.2% (-0.9%, 1.4%) |
| Laxatives; n (%) | 527 (2.6%) | 706 (3.0%) | -0.3% (-0.6%, -0.0%) | 396/2 8%) | 385 (2.7%) | 0.1% (-0.3%, 0.5%) |
| Number of distinct medications | SE7 (E.O70) | 7 0 0 (5.0 7.0) | 0.070 ( 0.070, 0.070) | 550 (E.570) | 305 (E.770) | 0.170 ( 0.070, 0.070) |
| mean (sd) | 13.21 (6.31) | 13.38 (6.58) | -0.17 (-0.29, -0.05) | 13.13 (6.41) | 13.23 (6.39) | -0.10 (-0.24, 0.05) |
| median [IQR] | 12.00 [9.00, 17.00] | 12.00 [9.00, 17.00] | - (-, -) | 12.00 [9.00, 16.00] | 12.00 [9.00, 17.00] | - (-, -) |
| min, max | 1.00,60.00 | 1.00, 62.00 | - (-, -) | 1.00,60.00 | 1.00,62.00 | - (-, -) |
| Number of office visits | 815 (616) | 8.32 (6.21) | 0.17 ( 0.20 , 0.05) | 8.05 (6.14) | 0.10 (5.03) | -0.05 (-0.19, 0.09) |
| mean (sd)median [IQR] | 7.00 [4.00,11.00] | 7.00 [4.00,11.00] | -0.17 (-0.28, -0.05)<br>- (-,-) | 6.00 [4.00, 10.00] | 8.10 (5.93)<br>7.00 [4.00,11.00] | -(-,-) |
| _min,max | 0.00,83.00 | 0.00,101.00 | - (-,-)<br> - (-,-) | 0.00,83.00 | 0.00,88.00 | - (-, -)<br>- (-, -) |
| Number of endocrinologist visits | 0.00,65.00 | 0.00,10100 | - (-,-) | 0.00,63.00 | 0.00,56.00 | - (-, -) |
| mean (sd) | 0.39 (1.24) | 0.38 (1.19) | 0.01 (-0.01, 0.04) | 0.38 (1.21)<br>0.00 [0.00, 0.00] | 0.38 (1.16) | -0.01 (-0.03, 0.02) |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) | 0.00 [0.00, 0.00] | 0.38 (1.16)<br>0.00 [0.00, 0.00] | - (-, -) |
| min, max | 0.00,30.00 | 0.00,25.00 | - (-, -) | 0.00,21.00 | 0.00,22.00 | - (-, -) |
| Number of cardiologist visits | | | | | | |
| _mean (sd) | 1.01 (2.72) | 0.83 (2.21) | 0.18 (0.13, 0.22) | 0.89 (2.53) | 0.89 (2.27) | 0.00 (-0.05, 0.06) |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | - (-, -)<br>- (-, -) | 0.00 [0.00,1.00] | 0.00 [0.00,1.00] | - (-, -)<br>- (-, -) |
| Number of internal/family medicine visits | 0.00,67.00 | 0.00,49.00 | - (-, -) | 0.00,67.00 | 0:00,44:00 | - (-, -) |
| mean (sd) | 4.94 (5.87) | 4.55 (5.48) | 0.39 (0.28, 0.50) | 4.67 (5.45) | 4.68 (5.96) | -0.01 (-0.14, 0.12) |
| median [IQR] | 4.00 [2.00, 6.00] | 3.00 [1.00, 6.00] | - (-, -) | 3.00 [1.00, 6.00] | 3.00 [1.00, 6.00] | - (-, -) |
| min, max | 0.00,216.00 | 0.00,364.00 | - (-, -) | 0.00,216.00 | 0.00, 364.00 | - (-, -) |
| Number of Electrocardiograms (ECG/EKG) | | | | | | |
| mean (sd) | 0.76 (1.46) | 0.66 (1.24) | 0.09 (0.07, 0.12) | 0.68 (1.35) | 0.69 (1.30) | -0.01 (-0.04, 0.02) |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | - (-, -) | 0.00 [0.00,1.00] | 0.00 [0.00,1.00] | - (-, -) |
| _min, max<br>Number of Echocardiograms | 0.00,28.00 | 0.00,24.00 | - (-, -) | 0.00,28.00 | 0.00,20.00 | - (-, -) |
| mean (sd) | 0.23 (0.67) | 0.19 (0.56) | 0.04 (0.03, 0.05) | 0.20 (0.62) | 0.20 (0.58) | -0.00 (-0.02, 0.01) |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-,-) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | -(-,-) |
| min, max | 0.00,12.00 | 0.00,11.00 | - (-, -) | 0.00,12.00 | 0.00,8.00 | - (-, -) |
| Out-of-pocket medication cost | | | | | | |
| mean (sd) | 525.68 (813.50) | 539.23 (1,028.23) | -13.55 (-30.82, 3.73) | 528.54 (827.61) | 534.96 (853.54) | -6.42 (-25.87,13.02) |
| median [IQR] | 318.00 [124.20, 672.49] | 296.03 [110.00, 670.00] | - (-, -) | 319.72 [119.28, 671.63] | 298.20 [112.10, 673.22] | - (-, -) |
| _min, max | -2,250.20,25,168.68 | -5,760.00,54,171.99 | - (-, -) | -553.97,25,168.68 | -5,760.00,20,191.25 | - (-, -) |
| Unique brand medicines<br>mean (sd) | 13.44 (6.49) | 13.60 (6.75) | -0.16 (-0.29, -0.04) | 13.34 (6.58) | 13.44 (6.57) | -0.10 (-0.25, 0.05) |
| mean (sd)<br>median [IQR] | 12.00 [9.00,17.00] | 12.00 [9.00,17.00] | -0.16 (-0.29, -0.04)<br>- (-, -) | 12.00 [9.00, 17.00] | 12.00 [9.00,17.00] | -0.10 (-0.25, 0.05)<br>- (-, -) |
| _min.max | 1.00,61.00 | 1.00.62.00 | - (-,-) | 1.00,61.00 | 1.00,62.00 | - (-, -)<br>- (-, -) |
| Unique generic medicines | | | | | | 117 |
| mean (sd) | 13.21 (6.31) | 13.38 (6.58) | -0.17 (-0.29, -0.05) | 13.13 (6.41) | 13.23 (6.39) | -0.10 (-0.24, 0.05) |
| median [IQR] | 12.00 [9.00, 17.00] | 12.00 [9.00,17.00] | - (-, -) | 12.00 [9.00, 16.00] | 12.00 [9.00, 17.00] | - (-, -) |
| min, max | 1.00,60.00 | 1.00, 62.00 | - (-, -) | 1.00, 60.00 | 1.00,62.00 | - (-, -) |
| Colonoscopy Sigmoidoscopy; n (%) | 1,996 (10.0%) | 2,592 (10.9%) | -0.9% (-1.5%, -0.3%) | 1,520 (10.6%) | 1,501 (10.5%) | 0.1% (-0.6%, 0.8%) |
| Flu Pneumococcal vaccine; n(%) Pap smear; n(%) | 6,142 (30.8%)<br>1.911 (9.6%) | 6,164 (25.9%)<br>3,024 (12.7%) | 4.9% (4.1%, 5.8%)<br>-3.1% (-3.7%, -2.5%) | 4,110 (28.6%)<br>1,561 (10.9%) | 4,081 (28.4%)<br>1,558 (10.9%) | 0.2% (-0.8%, 1.3%) |
| PSA test; n (%) | 4,103 (20.6%) | 5,004 (21.0%) | -0.4% (-1.2%, 0.3%) | 2,974 (20.7%) | 3,012 (21.0%) | -0.3% (-1.2%, 0.7%) |
| Fecal occult blood test; n (%) | 639 (3.2%) | 818 (3.4%) | -0.2% (-0.6%, 0.1%) | 466 (3.2%) | 488 (3.4%) | -0.2% (-0.6%, 0.3%) |
| Bone mineral density tests; n(%) | 616 (3.1%) | 814 (3.4%) | -0.3% (-0.7%, 0.0%) | 472 (3.3%) | 411 (2.9%) | 0.4% (0.0%, 0.8%) |
| Mammograms; n (%) | 4,755 (23.9%) | 6,520 (27.4%) | -3.5% (-4.4%, -2.7%) | 3.693 (25.7%) | 3,625 (25.2%) | 0.5% (-0.5%, 1.5%) |
| Telemedicine; n (%) | 5,769 (29.0%) | 6,961 (29.3%) | -0.3% (-1.2%, 0.5%) | 4,137 (28.8%) | 4,117 (28.7%) | 0.1% (-0.9%, 1.2%) |
| HbA1C tests | | 6,961 (29.3%) | -0.3% (-1.2%, 0.5%) | 4,137 (28.8%) | | |
| HbA1C tests<br>mean (sd) | 2.21 (1.44) | 6,961 (29.3%)<br>2.16 (1.42) | -0.3% (-1.2%, 0.5%)<br>0.05 (0.02, 0.07) | 4,137 (28.8%)<br>2.18 (1.41) | 2.19 (1.54) | -0.01 (-0.04, 0.03) |
| HbA1C tests _mean (sd) _median [IQR] | 2.21 (1.44)<br>2.00 [1.00, 3.00] | 6,961 (29.3%)<br>2.16 (1.42)<br>2.00 [1.00, 3.00] | -0.3% (-1.2%, 0.5%)<br>0.05 (0.02, 0.07)<br>- (-,-) | 4,137 (28.8%)<br>2.18 (1.41)<br>2.00 [1.00, 3.00] | 2.19 (1.54)<br>2.00 [1.00, 3.00] | -0.01 (-0.04, 0.03)<br>- (-, -) |
| HbAIC tests _mean(sd) _median(IQR) _min, max | 2.21 (1.44) | 6,961 (29.3%)<br>2.16 (1.42) | -0.3% (-1.2%, 0.5%)<br>0.05 (0.02, 0.07) | 4,137 (28.8%)<br>2.18 (1.41) | 2.19 (1.54) | -0.01 (-0.04, 0.03) |
| HbA1C tests _mean (sd) _median [IQR] | 2.21 (1.44)<br>2.00 [1.00, 3.00] | 6,961 (29.3%)<br>2.16 (1.42)<br>2.00 [1.00, 3.00] | -0.3% (-1.2%, 0.5%)<br>0.05 (0.02, 0.07)<br>- (-,-) | 4,137 (28.8%)<br>2.18 (1.41)<br>2.00 [1.00, 3.00] | 2.19 (1.54)<br>2.00 [1.00, 3.00] | -0.01 (-0.04, 0.03)<br>- (-, -) |
| HbAIC testsmean [sd]median [lQR]min, max Lipid panels | 2.21 (1.44)<br>2.00 (1.00, 3.00)<br>0.00, 41.00<br>1.48 (1.48)<br>1.00 (1.00, 2.00) | 6,961 (29.3%) 2.16 (1.42) 2.00 [1.00, 3.00] 0.00, 66.00 1.58 (1.18) 1.00 [1.00, 2.00] | -0.3% (-1.2%, 0.5%)<br>0.05 (0.02, 0.07)<br>- (-, -)<br>- (-, -) | 4.137 (28.8%) 2.18 (1.41) 2.00 [1.00, 3.00] 0.00, 41.00 1.51 (1.21) 1.00 [1.00, 2.00] | 2.19(1.54)<br>2.00 [1.00, 3.00]<br>0.00, 66.00<br>1.53 (1.20)<br>1.00 [1.00, 2.00] | -0.01 (-0.04, 0.03)<br>- (-, -)<br>- (-, -) |
| HbAIC testsmean [sd]median [lQR]min_max | 2.21(1.44)<br>2.00 [1.00, 3.00]<br>0.00, 41.00<br>1.48 (1.48) | 6,961 (29.3%) 2.16 (1.42) 2.00 [1.00, 3.00] 0.00, 66.00 1.58 (1.18) | -0.3% (-12%, 0.5%)<br>0.05 (0.02, 0.07)<br>- (-,-)<br>- (-,-)<br>-0.09 (-0.12, -0.07) | 4,137 (28.8%) 2.18 (1.41) 2.00 [1.00, 3.00] 0.00, 41.00 1.51 (1.21) | 2.19 (1.54)<br>2.00 [1.00, 3.00]<br>0.00, 66.00 | -0.01 (-0.04, 0.03)<br>-(-,-)<br>-(-,-)<br>-0.02 (-0.05, 0.01) |
| HBAIC testsmean (sd)median (lQR)min_max | 2.21 (1.44)<br>2.00 [1.00, 3.00]<br>0.00, 41.00<br>1.48 (1.48)<br>1.00 [1.00, 2.00]<br>0.00, 126.00 | 6,961 (29.3%) 2.16 (1.42) 2.00 (1.00, 3.00) 0.00, 66.00 1.58 (1.18) 1.00 (1.00, 2.00) 0.00, 30.00 | -0.3% (-12%, 0.5%)<br>0.05 (0.02, 0.07)<br>-(-,-)<br>-(-,-)<br>-0.09 (-0.12, -0.07)<br>-(-,-) | 4.137 (28.8%) 2.18 (1.41) 2.00 [1.00, 3.00] 0.00, 41.00 1.51 (1.21) 1.00 [1.00, 2.00] 0.00, 31.00 | 2.19 (1.54)<br>2.00 [1.00, 3.00]<br>0.00, 66.00<br>1.53 (1.20)<br>1.00 [1.00, 2.00]<br>0.00, 30.00 | -0.01 (-0.04, 0.03)<br>-(·,-)<br>-(·,-)<br>-0.02 (-0.05, 0.01)<br>-(·,-) |
| HbAIC testsmean (sd)median (lQR)min_max Lipid panelsmean (sd)median (lQR)min_max Creatinine testsmean (sd) | 2.21 (1.44)<br>2.00 [1.00, 3.00]<br>0.00, 41.00<br>1.48 (1.48)<br>1.00 [1.00, 2.00]<br>0.00, 126.00<br>0.04 (0.34) | 6,961 (29.3%) 216(1.42) 2.00 [1.00, 3.00] 0.00, 66.00 1.58 (1.18) 1.00 [1.00, 2.00] 0.00, 3.0.00 0.03 (0.25) | -0.3% (-12%, 0.5%)<br>0.05 (0.02, 0.07)<br>-(-,-)<br>-(-,-)<br>-0.09 (-0.12, -0.07)<br>-(-,-)<br>-(-,-)<br>-(-,-) | 4137 (28.8%) 2.18 (1.41) 2.00 (1.00, 3.00) 0.00, 41.00 1.51 (1.21) 1.00 (1.00, 2.00) 0.00, 31.00 0.03 (0.23) | 2.19(1.54)<br>2.00 [1.00,3.00]<br>0.00,66.00<br>1.53 (1.20)<br>1.00 [1.00,2.00]<br>0.00,30.00 | -0.01(-0.04,0.03)<br>-(·,·)<br>-(·,·)<br>-0.02(-0.05,0.01)<br>-(·,·)<br>-(·,·)<br>-0.01(-0.01,0.00) |
| HBAIC testsmean (sd)median (lQR)min_max | 221(1.44)<br>2.00 [1.00, 3.00]<br>0.00, 41.00<br>1.48 [1.48)<br>1.00 [1.00, 2.00]<br>0.00, 126.00<br>0.04 [0.34]<br>0.00 [0.00, 0.00] | 6,961 (29.3%) 216(1.42) 2.00 [1.00, 3.00] 0.00, 66.00 1.58(1.18) 1.00 [1.00, 2.00] 0.00, 30.00 0.03(0.25) 0.001, 0.001 | -0.3% (-12%, 0.5%) 0.05 (0.02, 0.07) -(-,-) | 4.137 (28.8%) 2.18(1.41) 2.00 (1.00, 3.00) 0.00, 41.00 1.51 (1.21) 1.00 (1.00, 2.00) 0.00, 31.00 0.03 (0.23) 0.00 (0.00, 0.00) | 219 (1.54)<br>2.00 (1.00, 3.00]<br>0.00, 66.00<br>1.53 (1.20)<br>1.00 (1.00, 2.00]<br>0.00, 3.000<br>0.03 (0.28)<br>0.00 (1.00, 0.00] | -0.01(-0.04, 0.03)<br>-(-,-)<br>-(-,-)<br>-0.02(-0.05, 0.01)<br>-(-,-)<br>-(-,-)<br>-0.01(-0.01, 0.00) |
| HBAIC testsmean [sd]median [lQR]min_max | 2.21 (1.44)<br>2.00 [1.00, 3.00]<br>0.00, 41.00<br>1.48 (1.48)<br>1.00 [1.00, 2.00]<br>0.00, 126.00<br>0.04 (0.34) | 6,961 (29.3%) 216(1.42) 2.00 [1.00, 3.00] 0.00, 66.00 1.58 (1.18) 1.00 [1.00, 2.00] 0.00, 3.0.00 0.03 (0.25) | -0.3% (-12%, 0.5%)<br>0.05 (0.02, 0.07)<br>-(-,-)<br>-(-,-)<br>-0.09 (-0.12, -0.07)<br>-(-,-)<br>-(-,-)<br>-(-,-) | 4137 (28.8%) 2.18 (1.41) 2.00 (1.00, 3.00) 0.00, 41.00 1.51 (1.21) 1.00 (1.00, 2.00) 0.00, 31.00 0.03 (0.23) | 2.19(1.54)<br>2.00 [1.00,3.00]<br>0.00,66.00<br>1.53 (1.20)<br>1.00 [1.00,2.00]<br>0.00,30.00 | -0.01(-0.04,0.03)<br>-(·,·)<br>-(·,·)<br>-0.02(-0.05,0.01)<br>-(·,·)<br>-(·,·)<br>-0.01(-0.01,0.00) |
| HbAIC testsmean [sd]median [lQR]min_max | 221(1.44)<br>2.00 [1.00, 3.00]<br>0.00, 410.00<br>1.48 [1.48]<br>1.00 [1.00, 2.00]<br>0.00, 126.00<br>0.04 (0.34)<br>0.00 [0.00, 0.00]<br>0.00, 230.00<br>0.12 (0.91) | 6,961 (29.3%) 2.16(1.42) 2.00 (1.00,3.00) 0.00,6600 1.58 (1.18) 1.00 (1.00,2.00) 0.00,3.000 0.03 (0.25) 0.00 (1.00,0.00) 0.00,1.000 0.00 (1.00) 0.00 (1.00) | -0.3% (-12%, 0.5%) 0.05 (0.02, 0.07) -(-,-) | 4.137 (2.83%) 2.18 (1.41) 2.00 (1.00,3.00) 0.00,41.00 1.51 (1.21) 1.00 (1.00,2.00) 0.00,31.00 0.03 (0.23) 0.00 (0.00,0.00) 0.00,6.00 0.00,6.00 0.00,6.00 0.00,6.00 0.00,6.00 0.00,6.00 | 219(1.54)<br>2.00 (1.00, 3.00)<br>0.00, 66.00<br>153 (1.20)<br>1.00 (1.00, 2.00)<br>0.00, 30.00<br>0.03 (0.28)<br>0.00 (0.00, 0.00)<br>0.00, 10.00<br>0.01 (0.00, 0.00) | -0.01(-0.04, 0.03)<br>-(-,-)<br>-(-,-)<br>-0.02(-0.05, 0.01)<br>-(-,-)<br>-(-,-)<br>-0.01(-0.01, 0.00) |
| HBAIC testsmean (sd)median [IQR]min max | 221(1.44) 2.00 (1.00, 3.00) 0.00, 41.00 1.48 (1.48) 1.00 (1.00, 2.00) 0.00, 126.00 0.04 (0.34) 0.00 (0.00, 0.00) 0.02 (2.91) 0.02 (0.91) 0.00 (0.00, 0.00) | 6.961 (29.3%) 2.16(1.42) 2.00 (1.00, 3.00) 0.00, 66.00 1.58 (1.18) 1.00 (1.00, 2.00) 0.00, 3.0.00 0.00 (1.00, 0.00) 0.00 (1.00, 0.00) 0.00 (1.00, 0.00) 0.00 (1.00, 0.00) 0.00 (1.00, 0.00) | 0.3% (-1.2%, 0.5%) 0.05 (0.02, 0.07) ·(·,·) ·0.09 (-0.12, -0.07) ·(·,·) ·(·,·) 0.01 (0.00, 0.02) ·(·,·) ·(·,·) | 4.137 (28.8%) 2.18 (1.41) 2.00 (1.00, 3.00) 0.00, 41.00 1.51 (1.21) 1.00 (1.00, 2.00) 0.00, 31.00 0.00 (2.30) 0.00 (0.00, 0.00) 0.00 (0.00, 0.00) 0.00 (0.00, 0.00) 0.00 (0.00, 0.00) | 219(1.54)<br>2.00 (1.00, 3.00)<br>0.00, 66.00<br>1.53 (1.20)<br>1.00 (1.00, 2.00)<br>0.00, 3.000<br>0.03 (0.28)<br>0.00 (0.00, 0.00)<br>0.01 (0.67)<br>0.00 (0.00, 0.00) | -0.01(-0.04, 0.03)<br>-(-,-) |
| HbAIC testsmean [sd]median [lQR]min max Lipid panelsmean [sd]median [lQR]min max Crestrine testsmean [sd]median [lQR]median [lQR]min max Natriuretic peptide testsmean [sd]median [lQR]median [lQR]median [lQR]median [lQR]median [lQR]median [lQR]median [lQR]median [lQR]min max | 221(1.44)<br>2.00 [1.00, 3.00]<br>0.00, 410.00<br>1.48 [1.48]<br>1.00 [1.00, 2.00]<br>0.00, 126.00<br>0.04 (0.34)<br>0.00 [0.00, 0.00]<br>0.00, 230.00<br>0.12 (0.91) | 6,961 (29.3%) 2.16(1.42) 2.00 (1.00,3.00) 0.00,6600 1.58 (1.18) 1.00 (1.00,2.00) 0.00,3.000 0.03 (0.25) 0.00 (1.00,0.00) 0.00,1.000 0.00 (1.00) 0.00 (1.00) | 0.3% (12%, 0.5%) 0.05(0.02,0.07) -(-,-) | 4.137 (2.83%) 2.18 (1.41) 2.00 (1.00,3.00) 0.00,41.00 1.51 (1.21) 1.00 (1.00,2.00) 0.00,31.00 0.03 (0.23) 0.00 (0.00,0.00) 0.00,6.00 0.00,6.00 0.00,6.00 0.00,6.00 0.00,6.00 0.00,6.00 | 219(1.54)<br>2.00 (1.00, 3.00)<br>0.00, 66.00<br>153 (1.20)<br>1.00 (1.00, 2.00)<br>0.00, 30.00<br>0.03 (0.28)<br>0.00 (0.00, 0.00)<br>0.00, 10.00<br>0.01 (0.00, 0.00) | -0.01(-0.04,0.03)<br>-(-,-)<br>-(-,-)<br>-(-,0.02(-0.05,0.01)<br>-(-,-) |
| HbAIC testsmean (sd)median [lQR]min_max | 221(1.44) 2.00 (1.00, 3.00) 0.00, 41.00 1.48 (1.48) 1.00 (1.00, 2.00) 0.00, 12.600 0.04 (0.34) 0.00 (0.00, 0.00) 0.00, 2.300 0.12 (0.91) 0.00 (0.00, 0.00) 0.00 (0.00, 0.00) 0.00 (0.00, 0.00) 0.00 (0.00, 0.00) | 6.961 (29.3%) 2.16(1.42) 2.00 [1.00, 3.00] 0.00, 66.00 1.58 (1.18) 1.00 [1.00, 2.00] 0.00, 30.00 0.00 (0.00, 0.00] | 0.3% (12%, 0.5%) 0.05 (0.02, 0.07) -(-,-) | 4.137 (28.8%) 2.18 (1.41) 2.00 (1.00, 3.00) 0.00, 41.00 1.51 (1.21) 1.00 (1.00, 2.00) 0.00, 31.00 0.00 (3.00, 0.00) 0.00 (0.00, 0.00) | 219(1.54) 2.00 (1.00, 3.00) 0.00, 6.60 0 1.53 (1.20) 1.00 (1.00, 2.00) 0.00, 30.00 0.03 (0.28) 0.00 (1.00, 0.00) 0.00 (1.00) 0.01 (0.07) 0.00 (1.00) 0.00 (1.00) 0.00 (1.00) 0.00 (1.00) | -0.01(-0.04,0.03) -(-,-) |
| HBAIC testsmean [sd]median [lQR]min max Lipid panelsmean [sd]median [lQR]min max Crestrine testsmean [sd]median [lQR]min max Natriuretic peptid testsmean [sd]median [lQR]median [lQR]median [lQR]median [lQR]median [lQR]median [lQR]median [lQR]median [lQR]min max | 221(1.44) 2.00 [1.00, 3.00] 0.00, 410 0 1.48 (1.48) 1.00 [1.00, 2.00] 0.00, 1250 0 0.04 (0.34) 0.00 (0.00, 0.00) 0.00, 230 0 0.12 (0.91) 0.00 (0.00, 0.00) 0.00, 4.00 0 0.00 0 0.00 | 6,961 (29.3%) 2.16 (1.42) 2.00 (1.00, 3.00] 0.00, 6600 1.58 (1.18) 1.00 (1.00, 2.00] 0.00, 3.000 0.03 (0.25) 0.00 (1.00, 0.00] 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 0.00, 2.800 0.89 (1.58) | 0.3% (-1.2%, 0.5%) 0.05 (0.02, 0.07) -(-,-) | 4.137 (28.8%) 2.18 (1.41) 2.00 (1.00, 3.00) 0.00, 41.00 1.51 (1.21) 1.00 (1.00, 2.00) 0.00, 31.00 0.03 (0.23) 0.00 (1.00, 0.00) 0.00, 6.00 0.00 (1.00, 0.00) 0.00 (1.00, 0.00) 0.00, 6.00 0 | 219(1.54)<br>2.00 (1.00, 3.00)<br>0.00, 66.00<br>153 (1.20)<br>1.00 (1.00, 2.00)<br>0.00, 30.00<br>0.03 (0.28)<br>0.00 (1.00, 0.00)<br>0.00, 10.00<br>0.01 (0.00, 0.00)<br>0.01 (0.00, 0.00)<br>0.00, 2.000<br>0.000, 2.000<br>0.0000, 2.000<br>0.0000<br>0.00000, 2.000<br>0.0000<br>0.0000<br>0.0000<br>0.0000<br>0.0000<br>0.0000<br>0.000 | 0.01(0.04,0.03) -(c,-) -(c,-) -(0.02(-0.05,0.01) -(c,-) -(c,-) -(0.01(-0.01,0.00) -(c,-) -(c,-) -(0.00(-0.02,0.01) -(c,-) |
| HBAIC testsmean (sd)median [lQR]min maxlipid panelsmean (sd)median [lQR]min max | 221(1.44) 2.00 (1.00, 3.00) 0.00, 41.00 1.48 (1.48) 1.00 (1.00, 2.00) 0.00, 126.00 0.00, 126.00 0.00 (1.00, 0.00) | 6.961 (29.3%) 2.16(1.42) 2.00 [1.00, 3.00] 0.00, 65.00 1.58 (1.18) 1.00 [1.00, 2.00] 0.00, 3.0.00 0.00 (0.00, 0.00] 0.89 (1.58) 0.00 (0.00, 1.00] | 0.3% (1.2%, 0.5%) 0.05 (0.02, 0.07) -(-,-) | 4.137 (28.8%) 2.18 (1.41) 2.00 (1.00, 3.00] 0.00, 41.00 1.51 (1.21) 1.00 (1.00, 2.00] 0.00, 31.00 0.00 (3.00, 0.00] 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 0.00 (3.00, 0.00] | 219(1.54) 2.00 (1.00, 3.00) 0.00, 66.00 1.53 (1.20) 1.00 (1.00, 2.00) 0.00, 30.00 0.03 (0.28) 0.00 (1.00, 0.00) 0.00, 1.00, 0.00) 0.00 (1.00, 0.00) 0.00 (1.58) 0.00 (1.00, 1.00) | -0.01(-0.04,0.03) -(-,-) -(-,-) -(-,-) -0.02(-0.05,0.01) -(-,-) |
| HbAIC tests | 221(1.44) 2.00 [1.00, 3.00] 0.00, 410 0 1.48 (1.48) 1.00 [1.00, 2.00] 0.00, 1250 0 0.04 (0.34) 0.00 (0.00, 0.00) 0.00, 230 0 0.12 (0.91) 0.00 (0.00, 0.00) 0.00, 4.00 0 0.00 0 0.00 | 6,961 (29.3%) 2.16 (1.42) 2.00 (1.00, 3.00] 0.00, 6600 1.58 (1.18) 1.00 (1.00, 2.00] 0.00, 3.000 0.03 (0.25) 0.00 (1.00, 0.00] 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 0.00, 2.800 0.89 (1.58) | 0.3% (-1.2%, 0.5%) 0.05 (0.02, 0.07) -(-,-) | 4.137 (28.8%) 2.18 (1.41) 2.00 (1.00, 3.00) 0.00, 41.00 1.51 (1.21) 1.00 (1.00, 2.00) 0.00, 31.00 0.03 (0.23) 0.00 (1.00, 0.00) 0.00, 6.00 0.00 (1.00, 0.00) 0.00 (1.00, 0.00) 0.00, 6.00 0 | 219(1.54)<br>2.00 (1.00, 3.00)<br>0.00, 66.00<br>153 (1.20)<br>1.00 (1.00, 2.00)<br>0.00, 30.00<br>0.03 (0.28)<br>0.00 (1.00, 0.00)<br>0.00, 10.00<br>0.01 (0.00, 0.00)<br>0.01 (0.00, 0.00)<br>0.00, 2.000<br>0.000, 2.000<br>0.0000, 2.000<br>0.0000<br>0.00000, 2.000<br>0.0000<br>0.0000<br>0.0000<br>0.0000<br>0.0000<br>0.0000<br>0.000 | 0.01(0.04,0.03) -(c,-) -(c,-) -(0.02(-0.05,0.01) -(c,-) -(c,-) -(0.01(-0.01,0.00) -(c,-) -(c,-) -(0.00(-0.02,0.01) -(c,-) |
| HBAIC testsmean (sd)median [lQR]min maxlipid panelsmean (sd)median [lQR]min max | 221(1.44) 2.00 (1.00, 3.00) 0.00, 41.00 1.48 (1.48) 1.00 (1.00, 2.00) 0.00, 126.00 0.00, 126.00 0.00 (1.00, 0.00) | 6.961 (29.3%) 2.16(1.42) 2.00 [1.00, 3.00] 0.00, 65.00 1.58 (1.18) 1.00 [1.00, 2.00] 0.00, 3.0.00 0.00 (0.00, 0.00] 0.89 (1.58) 0.00 (0.00, 1.00] | 0.3% (1.2%, 0.5%) 0.05 (0.02, 0.07) -(-,-) | 4.137 (28.8%) 2.18 (1.41) 2.00 [1.00.300] 0.00, 41.00 1.51 (1.21) 1.00 [1.00, 2.00] 0.00, 31.00 0.00 (3.00) 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 0.00 (47.00 0.86 (18.3) 0.00 (9.00, 1.00] | 219(1.54) 2.00 (1.00, 3.00) 0.00, 66.00 1.53 (1.20) 1.00 (1.00, 2.00) 0.00, 30.00 0.03 (0.28) 0.00 (1.00, 0.00) 0.00, 1.00, 0.00) 0.00 (1.00, 0.00) 0.00 (1.58) 0.00 (1.00, 1.00) | -0.01(-0.04,0.03) -(-,-) -(-,-) -(-,-) -0.02(-0.05,0.01) -(-,-) |
| HBAIC testsmean (sd)median [lQR]min maxlipid panelsmean (sd)median [lQR]min max | 221(1.44) 2.00 (1.00, 3.00) 0.00, 41.00 1.48 (1.48) 1.00 (1.00, 2.00) 0.00, 126.00 0.00 (1.00, 3.4) 0.00 (1.00, 0.00) 0.00 (2.300 0.12 (0.91) 0.00 (1.00, 0.00) | 6.961 (29.3%) 2.16(1.42) 2.00 (1.00, 3.00) 0.00, 66.00 1.58 (1.18) 1.00 (1.00, 2.00) 0.00, 3.0.00 0.00 (1.00, 0.00) 0.00 (1.00, 1.00) 0.00 (1.00, 1.00) | 0.3% (12%, 0.5%) 0.05 (0.02, 0.07) -(-,-) | 4.137 (28.8%) 2.18 (1.41) 2.00 [1.00.300] 0.00, 41.00 1.51 (1.21) 1.00 [1.00, 2.00] 0.00, 31.00 0.00 (3.00) 0.00 (0.00, 0.00] 1.00 (1.64) 1.00 (1.64) 1.00 (1.64) | 219(1.54) 2.00 (1.00, 3.00) 0.00, 66.00 1.53 (1.20) 1.00 (1.00, 2.00) 0.00, 30.00 0.00, 30.00 0.00 (1.00, 2.00) 0.00 (1.00, 2.00) 0.00 (1.00, 0.00) | -0.01(-0.04, 0.03) -(-,-) |
| HbAIC tests | 221(1.44) 2.00 [1.00, 3.00] 0.00, 410 0 1.48 (1.48) 1.00 [1.00, 2.00] 0.01, 250 0 0.01, 250 0 0.04 (0.34) 0.00 (0.00, 0.00) 0.00, 230 0 0.12 (0.91) 0.00 (0.00, 0.00) 0.00, 4.00 0 0.00, 9.10 0 0.00, 9.10 0 117 (1.81) | 6,961 (29.3%) 216(1.42) 2.06 (1.00, 3.00) 0.00, 6600 1.58 (1.8) 1.00 (1.00, 2.00) 0.00, 3.000 0.00 (3.025) 0.00 (0.00, 0.00) | 0.3% (-1.2%, 0.5%) 0.05 (0.02, 0.07) -(-,-) | 4.137 (28.8%) 2.18 (1.41) 2.00 (1.00, 3.00) 0.00, 41.00 1.51 (1.21) 1.00 (1.00, 2.00) 0.00, 31.00 0.03 (0.23) 0.00 (0.00, 0.00) 0.00, 0.00 0.00 (0.00, 0.00) 0.00 (0.00, 0.00) 0.00, 0.00 0.00 (0.00, 0.00) 0.00, 6.00 0.00, | 219(1.54)<br>2.00 (1.00, 3.00)<br>0.00, 6600<br>153 (1.20)<br>1.00 (1.00, 2.00)<br>0.00, 3000<br>0.03 (0.28)<br>0.00 (1.00, 0.00)<br>0.00, 1.000<br>0.01 (1.067)<br>0.00 (1.00, 0.00)<br>0.00, 2.000<br>0.00, 3.000<br>0.000, 3.000<br>0.0000, 3.000<br>0.00000, 3.000<br>0.0000, 3.000<br>0.0000, 3.000<br>0 | 0.01(0.04,0.03) -(x-) -( |
| HBAIC testsmean (sd)median [lQR]min max Lipid panelsmean (sd)median [lQR]min max | 221(1.44) 2.00 (1.00, 3.00) 0.00, 4100 1.48 (1.48) 1.00 (1.00, 2.00) 0.00, 126.00 0.00, 126.00 0.00 (1.00, 2.00) 0.00 (1.00, 2.00) 0.00 (1.00, 2.00) 0.00 (1.00, 0.00) | 6.961 (29.3%) 2.16(1.42) 2.00 (1.00, 3.00) 0.00, 66.00 1.58 (1.18) 1.00 (1.00, 2.00) 0.00, 3.0.00 0.00 (2.5) 0.00 (0.00, 0.00) 0.00 (0.00, 1.00) 0.00 (0.00, 1.00) 0.00 (0.00, 1.00) 0.00 (0.00, 0.00) | 0.3% (12%, 0.5%) 0.05 (0.02, 0.07) -(-,-) | 4.137 (28.8%) 2.18 (1.41) 2.00 (1.00.300] 0.00, 41.00 1.51 (1.21) 1.00 (1.00, 2.00] 0.00, 31.00 0.00 (3.00) 0.00 (0.00, 0.00] | 219(1.54) 2.00 (1.00, 3.00) 0.00, 66.00 1.53 (1.20) 1.00 (1.00, 2.00) 0.00, 30.00 0.00, 30 | -0.01(-0.04,0.03) -(-,-) -(-,-) -(-,-) -0.02(-0.05,0.01) -(-,-) |
| HbAIC tests | 221(1.44) 2.00 [1.00, 3.00] 0.00, 410 0 1.48 (1.48) 1.00 [1.00, 2.00] 0.00, 1250 0 0.01 (2.00) 0.01 (2.00) 0.00, 1250 0 0.01 (2.00) 0.00, 120 0 0.00, 120 0 0.00, 120 0 0.00, 17 (1.81) 1.00 [0.00, 2.00] 0.00, 1.00 0 1.17 (1.81) 1.00 [0.00, 2.00] 2.20 (1.50 0 0.15 (0.04) | 6,961 (29.3%) 2.16(1.42) 2.00 (1.00, 3.00) 0.00, 66.00 1.58 (1.18) 1.00 (1.00, 2.00) 0.00, 3.00.0 0.00 (3.00.0 0.00 (3.00. | 0.3% (-1.2%, 0.5%) 0.05 (0.02, 0.07) -() | 4.137 (28.8%) 2.18 (1.41) 2.200 (1.00, 3.00) 0.00, 41.00 1.51 (1.21) 1.00 (1.00, 2.00) 0.00, 31.00 0.03 (0.23) 0.00 (0.00, 0.00) 0.00, 0.00 0.00 (0.00, 0.00) 0.00 (0.00, 0.00) 0.00, 0.00 0.00 (0.00, 0.00) 0.00, 4.00 0.00 | 219(1.54) 2.00 (1.00, 3.00) 0.00, 66.00 1.53 (1.20) 1.00 (1.00, 2.00) 0.00, 3.00 0.00, | 0.01(0.04,0.03) -(-,-) |
| HBAIC testsmean (sd)median [lQR]min max Lipid panelsmean (sd)median [lQR]min max Creatine testsmean (sd)median [lQR]min max Natriuretic peptide testsmean (sd)median [lQR]min max Natriuretic peptide testsmean (sd)median [lQR]min max Urine testsmean (sd)min max Combined comorbidity scoremean (sd)min maxmedian [lQR]min maxmedian [lQR] | 221(1.44) 2.00 (1.00, 3.00) 0.00, 41.00 1.48 (1.48) 1.00 (1.00, 2.00) 0.00, 126.00 0.00, 126.00 0.00 (1.00, 2.00) 0.00 (1.00, 2.00) 0.00 (1.00, 2.00) 0.00 (1.00, 2.00) 0.00 (1.00, 0.00) | 6,961 (29.3%) 216(1.42) 2.00 [1.00, 3.00] 0.00, 650.0 1.58 (1.18) 1.00 [1.00, 2.00] 0.00, 3.0.0 0.03 (0.25) 0.00 (0.00, 0.00] 0.00 (0.00, 1.00] 0.00 (0.00, 1.00] 0.00 (0.00, 0.00] | 0.3% (1.2%, 0.5%) 0.05 (0.02, 0.07) -(-,-) | 4.137 (28.8%) 2.18 (1.41) 2.00 (1.00.300] 0.00, 41.00 1.51 (1.21) 1.00 (1.00.2.00] 0.00, 31.00 0.00 (2.30) 0.00 (0.00) | 219(1.54) 2.09 (1.00, 3.00) 0.00, 66.00 1.53 (1.20) 1.00 (1.00, 2.00) 0.00, 30.00 0.00, 30 | -0.01(-0.04,0.03) -(-,-) |
| HbAIC testsmean [sd]median [lQR]min max Lipid panelsmean [sd]median [lQR]min max Creatrine testsmean [sd]median [lQR]min max Natriuretic peptide testsmean [sd]median [lQR]median [lQR]min max Urine testsmean [sd]median [lQR]median [lQR]min max | 221(1.44) 2.00 [1.00, 3.00] 0.00, 410 0 1.48 (1.48) 1.00 [1.00, 2.00] 0.00, 1250 0 0.01 (2.00) 0.01 (2.00) 0.00, 1250 0 0.01 (2.00) 0.00, 120 0 0.00, 120 0 0.00, 120 0 0.00, 17 (1.81) 1.00 [0.00, 2.00] 0.00, 1.00 0 1.17 (1.81) 1.00 [0.00, 2.00] 2.20 (1.50 0 0.15 (0.04) | 6,961 (29.3%) 2.16(1.42) 2.00 (1.00, 3.00) 0.00, 66.00 1.58 (1.18) 1.00 (1.00, 2.00) 0.00, 3.00.0 0.00 (3.00.0 0.00 (3.00. | 0.3% (-1.2%, 0.5%) 0.05 (0.02, 0.07) -() | 4.137 (28.8%) 2.18 (1.41) 2.200 (1.00, 3.00) 0.00, 41.00 1.51 (1.21) 1.00 (1.00, 2.00) 0.00, 31.00 0.03 (0.23) 0.00 (0.00, 0.00) 0.00, 0.00 0.00 (0.00, 0.00) 0.00 (0.00, 0.00) 0.00, 0.00 0.00 (0.00, 0.00) 0.00, 4.00 0.00 | 219(1.54) 2.00 (1.00, 3.00) 0.00, 66.00 1.53 (1.20) 1.00 (1.00, 2.00) 0.00, 3.00 0.00, | 0.01(0.04,0.03) -(-,-) |
| HbAIC testsmean (sd)median [lQR]min max Lipid panelsmean (sd)median [lQR]min max Creatine testsmean (sd)median [lQR]min max Creatine testsmean (sd)median [lQR]min max Natriuretic peptide testsmean (sd)median [lQR]min max Urine testsmean (sd)min max Urine testsmean (sd)min maxmedian [lQR]min maxmedian [lQR] | 221(1.44) 2.00 (1.00, 3.00) 0.00, 4100 1.48 (1.48) 1.00 (1.00, 2.00) 0.00, 126.00 0.00, 126.00 0.00 (2.00) 0.00, 2.300 0.12 (0.91) 0.00 (0.00, 0.00) 0.00, 7.00 0.00 (0.00, 1.00) | 6,961 (29.3%) 216(1.42) 2.00 [1.00, 3.00] 0.00, 650.0 1.58 (1.18) 1.00 [1.00, 2.00] 0.00, 3.0.0 0.03 (0.25) 0.00 (0.00, 0.00] 0.00 (0.00, 1.00] 0.00 (0.00, 1.00] 0.00 (0.00, 1.00] 0.00 (0.00, 1.00] 0.00 (0.00, 1.00] 0.00 (0.00, 0.00] | 0.3% (12%, 0.5%) 0.05 (0.02, 0.07) -(-,-) | 4.137 (28.8%) 2.18 (1.41) 2.00 (1.00.300] 0.00, 41.00 1.51 (1.21) 1.00 (1.00.2.00] 0.00, 31.00 0.00 (3.00) 0.00 (0.00, 0.00] | 219(1.54) 2.00 (1.00, 3.00) 0.00, 66.00 1.53 (1.20) 1.00 (1.00, 2.00) 0.00, 30.00 0.03 (0.28) 0.00 (1.00, 0.00) 0.00, 1.00 0.00 0.00, 1.00 0.00 0.00 0.00 0.00 0.00 0.00 0.00 | -0.01(-0.04,0.03) -(-,-) |
| HBAIC testsmean (sd)median [lQR]min max Lipid panelsmean (sd)median [lQR]min max Creatine testsmean (sd)median [lQR]min max Natriuretic peptide testsmean (sd)median [lQR]min max Natriuretic peptide testsmean (sd)median [lQR]min max Urine testsmean (sd)min max Combined comorbidity scoremean (sd)min maxmedian [lQR]min maxmore fleepitalizations | 221(1.44) 2.00 [1.00, 3.00] 0.00, 4100 1.48 (1.48) 1.00 [1.00, 2.00] 0.00, 12600 0.01 (2.00) 0.01 (2.00) 0.00, 12600 0.01 (2.00) 0.00, 1200 0.00, 1200 0.00, 1000 | 6,961 (29.3%) 2.16(1.42) 2.00 (1.00, 3.00) 0.00, 66.00 1.58 (1.8) 1.00 (1.00, 2.00) 0.00, 3.00.0 0.00, 3.00.0 0.00 (2.5) 0.00 (0.00, 0.00) | 0.3% (1.2%, 0.5%) 0.05 (0.02, 0.07) -(-,-) | 4.137 (28.8%) 2.18 (1.41) 2.20 (1.100, 3.00] 0.00, 410.0 1.51 (1.21) 1.00 (1.00, 2.00] 0.00, 3.10.0 0.00 (3.00) 0. | 219(1.54) 2.09 (1.00, 3.00) 0.00, 66.00 1.53 (1.20) 1.00 (1.00, 2.00) 0.00, 30.00 0.00, 30 | -0.01(-0.04,0.03) -(-,-) |
| HbAIC tests | 221(1.44) 2.00 [1.00, 3.00] 0.00, 410 0 1.48 (1.48) 1.00 [1.00, 2.00] 0.01, 2.00] | 6,961 (29.3%) 2.16(1.42) 2.00 (1.00, 3.00) 0.00, 66.00 1.58 (1.18) 1.00 (1.00, 2.00) 0.00, 3.00.0 0.00, 3.00.0 0.00 (2.50) | 0.3% (-1.2%, 0.5%) 0.05 (0.02, 0.07) -() | 4.137 (28.8%) 2.18 (1.41) 2.200 (1.00, 3.00) 0.00, 410.0 1.51 (1.21) 1.00 (1.00, 2.00) 0.00, 3.10.0 0.00 (3.00) | 219(1.54) 2.00 (1.00, 3.00) 0.00, 66.00 1.53 (1.20) 1.00 (1.00, 2.00) 0.00, 3.00 0.00 0.00, 3.00 0.00 0.00, 3.00 0.00 0.00 0.00 0.00 0.00 0.00 0.00 | 0.01(0.04,0.03) -(c,-) -(c,-) -(0.02(0.05,0.01) -(c,-) -(c,-) -(0.01(0.01,0.00) -(c,-) -(c,-) -(0.00(0.02,0.01) -(c,-) -(c,-) -(0.00(0.04,0.04) -(c,-) |
| HBAIC testsmean (sd)median [lQR]min max Lipid panelsmean (sd)median [lQR]min max Creatinine testsmean (sd)median [lQR]min max Natriuretic peptide testsmean (sd)median [lQR]min max Natriuretic peptide testsmean (sd)median [lQR]min max Urine testsmean (sd)min max Combined comorbidity scoremean (sd)min maxmedian [lQR]min maxmean (sd)median [lQR]min maxmean (sd)median [lQR]min maxmean (sd)median [lQR]min maxmean (sd)median [lQR]min maxmean (sd)median [lQR]min max | 221(1.44) 2.00 (1.00, 3.00) 0.00, 4100 1.48 (1.48) 1.00 (1.00, 2.00) 0.00, 126.00 0 | 6.96I (29.3%) 2.16(1.42) 2.00 [1.00, 3.00] 0.00, 65.00 1.58 (1.18) 1.00 [1.00, 2.00] 0.00, 3.0.00 0.00 (0.00, 0.00] 0.00 (0.00, 1.00] 0.00 (0.00, 1.00] 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 0.01 (0.00, 0.00] 0.01 (0.00, 0.00] 0.01 (0.00, 0.00] 0.01 (0.00, 0.00] 0.01 (0.00, 0.00] 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] | 0.3% (12%, 0.5%) 0.05 (0.02, 0.07) -(-,-) | 4.137 (28.8%) 2.18 (1.41) 2.00 (1.00.300] 0.00, 41.00 1.51 (1.21) 1.00 (1.00.2.00] 0.00, 31.00 0.03 (2.3) 0.03 (0.23) 0.03 (0.23) 0.03 (0.23) 0.00 (0.00, 0.00] | 219(1.54) 2.00 (1.00, 3.00) 0.00, 66.00 1.53 (1.20) 1.00 (1.00, 2.00] 0.00, 3.00 0.00, | -0.01(-0.04,0.03) -(-,-) -(-,-) -(-,0.02(-0.05,0.01) -(-,-) -(-,- |
| HbAIC testsmean [sd]median [lQR]min max Lipid panelsmean [sd]median [lQR]min max Creatrine testsmean [sd]median [lQR]min max Natriuretic peptide testsmean [sd]median [lQR]min max Urine testsmean [sd]median [lQR]median [lQR]min max Urine testsmean [sd]median [lQR]median [lQR]min max Combined comorbidity scoremean [sd]median [lQR]median [lQR]min max Frailty Scoremean [sd]median [lQR]min max Number of Hospitalizationsmean [sd]median [lQR]median [lQR]min max Ary hospitalization within prior 92 - 365 days; n (%) | 221(1.44) 2.00 [1.00, 3.00] 0.00, 410 0 1.48 (1.48) 1.00 [1.00, 2.00] 0.01, 2.00] | 6,961 (29.3%) 2.16(1.42) 2.00 (1.00, 3.00) 0.00, 66.00 1.58 (1.18) 1.00 (1.00, 2.00) 0.00, 3.00.0 0.00, 3.00.0 0.00 (2.50) | 0.3% (-1.2%, 0.5%) 0.05 (0.02, 0.07) -() | 4.137 (28.8%) 2.18 (1.41) 2.200 (1.00, 3.00) 0.00, 410.0 1.51 (1.21) 1.00 (1.00, 2.00) 0.00, 3.10.0 0.00 (3.00) | 219(1.54) 2.00 (1.00, 3.00) 0.00, 66.00 1.53 (1.20) 1.00 (1.00, 2.00) 0.00, 3.00 0.00 0.00, 3.00 0.00 0.00, 3.00 0.00 0.00 0.00 0.00 0.00 0.00 0.00 | 0.01(0.04,0.03) -(c,-) -(c,-) -(0.02(0.05,0.01) -(c,-) -(c,-) -(0.01(0.01,0.00) -(c,-) -(c,-) -(0.00(0.02,0.01) -(c,-) -(c,-) -(0.00(0.04,0.04) -(c,-) |
| HBAIC testsmean (sd)median (lQR)min max Lipid panelsmean (sd)median (lQR)min max Creatinine testsmean (sd)median (lQR)min max Natrivetic poptide testsmean (sd)median (lQR)min max Natrivetic poptide testsmean (sd)median (lQR)min max Universitymedian (lQR)min maxmedian (lQR)min maxmaxmedian (lQR)min maxmay (sd)min may (sd)min ma | 221(1.44) 2.00 (1.00, 3.00) 0.00, 41.00 1.48 (1.48) 1.00 (1.00, 2.00) 0.00, 1.26 (0.00) 0.00, 1.26 (0.00) 0.00, 1.26 (0.00) 0.00, 1.20 (0.00) | 6.96I (29.3%) 2.16(1.42) 2.00 [1.00, 3.00] 0.00, 66.00 1.58 (1.18) 1.00 [1.00, 2.00] 0.00, 3.0.00 0.00 (0.00, 0.00] 0.01 (0.00, 0.00] 0.01 (0.00, 0.00] 0.01 (0.00, 0.00] 0.01 (0.00, 0.00] 0.01 (0.00, 0.00] 0.00 (0.00, 0.00] | 0.3% (12%, 0.5%) 0.05 (0.02, 0.07) -(-,-) -( | 4.137 (28.8%) 2.18 (1.41) 2.00 [1.00.300] 0.00, 41.00 1.51 (1.21) 1.00 [1.00, 2.00] 0.00, 31.00 0.00 (3.00) 0.00 (0.00, 0.00] | 219(1.54) 2.00 (1.00, 3.00) 0.00, 66.00 1.53 (1.20) 1.00 (1.00, 2.00] 0.00, 3.00 0.00, | -0.01(-0.04, 0.03) -(-,-) -(-,-) -(-,0.02(-0.05, 0.01) -(-,-) -(- |
| HbAIC tests | 221(1.44) 2.00 [1.00, 3.00] 0.00, 4100 1.48 (1.48) 1.00 [1.00, 2.00] 0.00, 12500 0.01 (2.00) 0.01 (2.00) 0.01 (2.00) 0.00, 2.00] 0.00, 2.00] 0.00, 2.00] 0.00, 2.00] 0.00, 2.00] 0.00, 4.00 0.00, 4.00 0.00, 4.00 0.00, 4.00 0.00, 4.00 0.00, 9.100 0.00, 9.100 0.00, 9.100 0.00, 9.100 0.00, 9.100 0.00, 9.100 0.00, 9.100 0.15 (0.00, 9.100) | 6,961 (29.3%) 2.16(1.42) 2.00 (1.00, 3.00) 0.00, 66.00 1.58 (1.18) 1.00 (1.00, 2.00) 0.00, 3.0.00 0.00, 3.0.00 0.00 (2.50) 0.00 (0.00, 0.00) 0.00 (2.700) 560 (2.4%) 1.239 (5.2%) | 0.3% (-12%, 0.5%) 0.05 (0.02, 0.07) -(-,-) | 4.137 (28.8%) 2.18 (1.41) 2.20 (1.100, 3.00] 0.00, 410.0 1.51 (1.21) 1.00 (1.00, 2.00] 0.00, 3.10.0 0.00 (3.10.0 0.00 (3.00.0 0.00 (3.0 | 219(1.54) 2.00 (1.00, 3.00) 0.00, 66.00 153 (1.20) 1.00 (1.00, 2.00) 0.00, 30.00 0.00, 30 | 0.01 (0.04, 0.03) -(-,-) -(-,- |
| HbAIC testsmean (sd)median (lQR)min max Lipid panelsmean (sd)median (lQR)min max Creatinine testsmean (sd)median (lQR)min max Natrivetic poptide testsmean (sd)median (lQR)min max Natrivetic poptide testsmean (sd)median (lQR)min max Universitymedian (lQR)min maxmedian (lQR)min maxmay = 1 days; n %6 Any hospitalization within prior 91 days; n %6 Any hospitalization within prior 92 - 365 days; n %6 | 221(1.44) 2.00 (1.00, 3.00) 0.00, 41.00 1.48 (1.48) 1.00 (1.00, 2.00) 0.00, 1.26 (0.00) 0.00, 1.26 (0.00) 0.00, 1.26 (0.00) 0.00, 1.20 (0.00) 0.20 (0.00) 0.20 (0.00) 0.20 (0.00) 0.30 (0. | 6.96I (29.3%) 2.16(1.42) 2.00 [1.00, 3.00] 0.00, 650.0 1.58 (1.18) 1.00 [1.00, 2.00] 0.00, 3.0.0 0.03 (0.25) 0.00 (0.00, 0.00] 0.00 (0.00, 1.00] 0.00 (0.00, 1.00] 0.00 (0.00, 1.00] 0.00 (0.00, 1.00] 0.01 (0.00, 0.00] 0.03 (1.58) 1.00 (0.00, 0.00] 0.01 (0.00, 0.00] 0.03 (1.00) 0.04 (0.04) 0.13 (0.12 (0.16) 0.04 (0.16) 0.13 (0.12 (0.16) 0.04 (0.16) 0.13 (0.12 (0.16) 0.13 (0.16) 0.13 (0.12 (0.16) 0.14 (0.04) 0.13 (0.12 (0.16) 0.14 (0.04) 0.13 (0.12 (0.16) 0.04 (0.16) 0.13 (0.12 (0.16) 0.04 (0.16) 0.13 (0.12 (0.16) 0.14 (0.04) | 0.3% (12%, 0.5%) 0.05 (0.02, 0.07) -(-,-) - | 4.137 (28.8%) 2.18 (1.41) 2.00 (1.00.300] 0.00, 41.00 1.51 (1.21) 1.00 (1.00.2.00] 0.00, 31.00 0.03 (2.3) 0.00 (0.00, 0.00] | 219(1.54) 2.00 (1.00, 3.00) 0.00, 66.00 1.53 (1.20) 1.00 (1.00, 2.00] 0.00, 3.00 0.00 0.00 0.00 0.00 0.00 0.00 0.00 | -0.01(-0.04, 0.03) -(-,-) -(-,-) -(-,0.02(-0.05, 0.01) -(-,-) -(- |
| HbAIC tests | 221(1.44) 2.00 [1.00, 3.00] 0.00, 4100 1.48 [1.48] 1.00 [1.00, 2.00] 0.01, 3.00] 0.01, 3.0 | 6,961 (29.3%) 2.16(1.42) 2.00 (1.00, 3.00) 0.00, 66.00 1.58 (1.18) 1.00 (1.00, 2.00) 0.00, 3.0.00 0.00, 3.0.00 0.00 (2.50) 0.00 (0.00, 0.00) 1.239 (5.2%) 2.2.133 (93.0%) 1.529 (6.4%) | 0.3% (12%, 0.5%) 0.05 (0.02, 0.07) -(-,-) | 4.137 (28.8%) 2.18 (1.41) 2.20 (1.100, 3.00] 0.00, 4100 1.51 (1.21) 1.00 (1.00, 2.00] 0.00, 3100 0.00 (3.100 0.00 (3.00) 0.00 (3.00) 0.00 (0.00, 0.00) 0.00 (0.00, 0.00) 0.00, 4.00 0.00 (0.00, 0.00) 0.00, 4.00 0.00 (0.00, 0.00) 0.00, 4.00 0.00 (0.00, 0.00) 0.00, 4.00 0.00 (1.00) 0.0 | 219(1.54) 2.00 (1.00, 3.00) 0.00, 66.00 1.53 (1.20) 1.00 (1.00, 2.00) 0.00, 3.00 0.00 0.00, 3.00 0. | 0.01 (0.04, 0.03) -(-,-) -(-,- |
| HbAIC tests | 221(1.44) 2.00 (1.00, 3.00) 0.00, 41.00 1.48 (1.48) 1.00 (1.00, 2.00) 0.00, 1.26 (0.00) 0.00, 1.26 (0.00) 0.00, 1.26 (0.00) 0.00, 1.20 (0.00) 0.20 (0.00) 0.20 (0.00) 0.20 (0.00) 0.30 (0. | 6.96I (29.3%) 2.16(1.42) 2.00 [1.00, 3.00] 0.00, 650.0 1.58 (1.18) 1.00 [1.00, 2.00] 0.00, 3.0.0 0.03 (0.25) 0.00 (0.00, 0.00] 0.00 (0.00, 1.00] 0.00 (0.00, 1.00] 0.00 (0.00, 1.00] 0.00 (0.00, 1.00] 0.01 (0.00, 0.00] 0.03 (1.58) 1.00 (0.00, 0.00] 0.01 (0.00, 0.00] 0.03 (1.00) 0.04 (0.04) 0.13 (0.12 (0.16) 0.04 (0.16) 0.13 (0.12 (0.16) 0.04 (0.16) 0.13 (0.12 (0.16) 0.13 (0.16) 0.13 (0.12 (0.16) 0.14 (0.04) 0.13 (0.12 (0.16) 0.14 (0.04) 0.13 (0.12 (0.16) 0.04 (0.16) 0.13 (0.12 (0.16) 0.04 (0.16) 0.13 (0.12 (0.16) 0.14 (0.04) | 0.3% (12%, 0.5%) 0.05 (0.02, 0.07) (;-) 0.01 (0.00, 0.02) (;-) -0.03 (0.01, 0.04) (;-) -0.04 (-0.07, -0.01) (;-) (;-) 0.24 (0.21, 0.27) (;-) 0.17 (0.00, 0.01) (;-) 1.5 (0.00, 0.01) (;-) 1.7 (1.53, 2.42) (;-) 1.97 (1.53, 2.42) (;-) 2.9% (1.5%, 2.5%) 2.9% (1.5%, 2.5%) 2.9% (2.5%, 2.5%) 2.9% (2.5%, 2.5%) 1.9% (0.5%, 2.5%) 1.9% (0.5%, 2.5%) 1.9% (0.5%, 2.5%) 1.9% (0.5%, 2.5%) | 4.137 (28.8%) 2.18 (1.41) 2.20 (1.100, 3.00] 0.00, 410.0 1.51 (1.21) 1.00 (1.00, 2.00] 0.00, 310.0 0.00, 310.0 0.00 (1.00, 2.00] 0.00 (1.00, 3.00) 0.00 (1.0 | 219(1.54) 2.00 (1.00, 3.00) 0.00, 66.00 1.53 (1.20) 1.00 (1.00, 2.00] 0.00, 3.00 0.00 0.00 0.00 0.00 0.00 0.00 0.00 | -0.01(-0.04, 0.03) -(-,-) -(-,-) -(-,0.02(-0.05, 0.01) -(-,-) -(- |
| HbAIC testsmean (sd)median (lQR)min max Lipid panelsmean (sd)median (lQR)min max Creatinine testsmean (sd)median (lQR)min max Natriuretic peptide testsmean (sd)median (lQR)min max Natriuretic peptide testsmean (sd)median (lQR)min max Urine testsmedian (lQR)min max Urine testsmedian (lQR)min max Fraity Scoremean (sd)median (lQR)min max Natriuretic peptide testsmedian (lQR)min max Natriuretic peptide testsmedian (lQR)min maxmedian ( | 221(1.44) 2.00 [1.00, 3.00] 0.00, 41.00 1.48 [1.48) 1.00 [1.00, 2.00] 0.00, 1.26 0.0 0.26 0.0 0.00, 1.26 0.0 0.27 0.0 0.27 0.0 0.00, 1.26 0.0 | 6,961 (29.3%) 2.16(1.42) 2.00 [1.00, 3.00] 0.00, 65.00 1.58 (1.18) 1.00 [1.00, 2.00] 0.00, 3.0.00 0.00 (0.00, 0.00] 0.01 (0.00, 0.00] 0.04 (0.04) 0.13 (0.12, 0.16) 0.04, 0.04 0.13 (0.12, 0.16) 0.04, 0.04 0.13 (0.12, 0.16) 0.04, 0.09 1.23 (0.27, 0.00) 1.24 (0.27, 0.00) 1.25 (0.27, 0 | 0.3% (12%, 0.5%) 0.05 (0.02, 0.07) -(-,-) - | 4.137 (28.8%) 2.18 (1.41) 2.00 [1.00.300] 0.00, 41.00 1.51 (1.21) 1.00 [1.00, 2.00] 0.00, 31.00 0.03 (0.23) 0.03 (0.23) 0.00 (0.00, 0.00] 0.00, 6.00 0.00 (0.00, 0.00] | 219 (1.54) 2.09 (1.00, 3.00) 0.00, 6.60 0 1.53 (1.20) 1.00 (1.00, 2.00] 0.00, 3.00 0 0.00, 3.00 | -0.01(-0.04, 0.03) -(-, -) -(- |
| HbAIC tests | 221 (1.44) 2.00 [1.00, 3.00] 0.00, 4100 1.48 (1.48) 1.00 [1.00, 2.00] 0.01, 3.00] 0.01, 3 | 6,961 (29.3%) 216(1.42) 2.00 [1.00, 3.00] 0.00, 66.00 1.58 (1.18) 1.00 [1.00, 2.00] 0.00, 3.0.00 0.00, 3.0.00 0.00 (0.00, 0.00] 0.14 (0.04) 0.13 (0.15 (0.00) 0.14 (0.04) 3.83 (20.05) 0.00 (0.00, 0.00] 0.00, 0.00 (0.00, 0.00) 1.25 (0.5%) 1.25 (0.5%) 1.25 (0.5%) 1.52 (6.4%) 3.07 (1.3%) 6.542 (27.5%) 164 (0.7%) 164 (0.7%) | 0.3% (12%, 0.5%) 0.05 (0.02, 0.07) (,-) 0.01 (0.00, 0.02) (,-) (,-) 0.03 (0.01, 0.04) (,-) (,-) -0.04 (-0.07, -0.01) (,-) (,-) 0.24 (0.21, 0.27) (,-) (,-) 1.57 0.01 (0.00, 0.01) (,-) 1.57 1.59 1.5 | 4.137 (28.8%) 2.18 (1.41) 2.20 (1.00, 3.00] 0.00, 4100 1.51 (1.21) 1.00 (1.00, 2.00] 0.00, 3100 0.00, 3100 0.00 (3.00) 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 0.00, 4.00 0.00 (0.00, 0.00] 0.00, 4.00 0.00 (0.00, 0.00] 0.00, 4.00 0.00, 5.05 4.41 (23.08) 0.90 (0.00, 0.00] 0.90, 73.80 0.90 (0.00, 0.00] 0.90, 74.80 0.90 (0.00, 0.00] 0.90, 74.80 0.90 (0.90, 0.00] 0.90, 74.80 0.90 (0.90, 0.90) 0.90, 74.90 0.90, 74 | 219 (1.54) 2.00 (1.00, 3.00) 0.00, 66.00 153 (1.20) 1.00 (1.00, 2.00) 0.00, 3.00 0.00 0.00, 3.00 0.00 0.00, 3.00 0.00 0.00 0.00 0.00 0.00 0.00 0.00 | 0.01 (0.04, 0.03) -(-,-) -(-,- |
| HbAIC testsmean (sd)median (lQR)min max Lipid panelsmean (sd)median (lQR)min max Creatinine testsmean (sd)median (lQR)min max Natriuretic peotide testsmean (sd)median (lQR)min max Urine testsmean (sd)median (lQR)min max Urine testsmedian (lQR)min max Urine testsmean (sd)median (lQR)min max Fraity Scoremean (sd)median (lQR)min max Natriuretic peotide testsmedian (lQR)min maxmedian (lQR)min maxmospitalization within prior 91 days; n (%) Any hospitalization within prior 92 - 365 days; n (%) Number of hospitalizations (0, 1, 2 or more)<br> | 221(1.44) 2.00 [1.00, 3.00] 0.00, 41.00 1.48 [1.48) 1.00 [1.00, 2.00] 0.00, 1.26 0.0 1.00 [1.00, 2.00] 0.00, 1.26 0.0 0.04 (0.34) 0.00 [1.00, 0.00] 0.00, 2.300 0.12 (0.91) 0.00 [1.00, 0.00] 0.00, 4.00 1.00 0.00, 0.00] 0.00, 4.00 1.00 0.00, 0.00 1.00 0.00, 4.00 1.00 0.00, 0.00 1.00 0.00, 1.00 0.00 0.00, 1.00 0.00 0.00, 1.00 0.00 0.00, 1. | 6,961 (29.3%) 216(1.42) 2.00 [1.00, 3.00] 0.00, 650.0 1.58 (1.18) 1.00 [1.00, 2.00] 0.03, 0.00 0.03, 0.00 0.03, 0.00 0.03, 0.00 0.00 [0.00, 0.00] 0.00 [0.00, 0.00] 0.00 [0.00, 0.00] 0.00 [0.00, 0.00] 0.00 [0.00, 0.00] 0.00, 280.0 0.89 (1.58) 0.00 [0.00, 1.00] 0.03, 34.00 0.93 (1.58) 1.00 [0.00, 2.00] 2.00, 14.00 1.00 [0.00, 2.00] 2.00, 14.00 1.35 [2.05] 0.04 (0.04) 1.35 [2.05] 0.00 [0.00, 0.00] 0.00, 2.700 560 (2.4%) 1.23 [9.2%) 1.25 [9.6%) 1.52 [9.6%] 1.52 [9.6%] | 0.3% (-12%, 0.5%) 0.05 (0.02, 0.07) (-, -) ( | 4.137 (28.8%) 2.18 (1.41) 2.00 (1.00.300] 0.00,410.0 1.51 (1.21) 1.00 (1.00.2.00] 0.00,310.0 0.00,310.0 0.00 (1.00.0.00] 0.00 (1.00.0.0.00] 0.00 (1.00.0.00] 0. | 219 (1.54) 2.09 (1.00, 3.00) 0.00, 66.00 1.53 (1.20) 1.00 (1.00, 2.00] 0.00, 3.00 0.00, | -0.01(-0.04, 0.03) -(-, -) -(- |
| HbAIC tests | 221(1.44) 2.00 [1.04) 2.00 [1.03.30] 0.00,4100 1.48 [1.48] 1.00 [1.00,2.00] 0.01,126.00 0.01,126.00 0.04 (0.34) 0.00 (1.00,0.00) 0.00,2.300 0.00,2.300 0.12 (0.91) 0.00 (1.00,0.00) 0.00,4.000 0.00,9.000 0.00,9.000 0.00,9.000 0.00,9.000 0.00,9.000 0.00,0.000 1.1444 (7.2%) 17.955 (90.1%) 124 (0.5%) 1848 (9.3%) 469 (2.14%) 69 (2.14%) 69 (2.14%) 69 (2.14%) 1357 (6.3%) 1357 (6.3%) 1357 (6.3%) | 6,961 (29.3%) 2.16(1.42) 2.00 [1.00, 3.00] 0.00, 66.00 1.58 (1.18) 1.00 [1.00, 2.00] 0.00, 3.0.00 0.00, 3.0.00 0.00 (0.00, 0.00] 0.14 (0.04) 3.83 (20.05) 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 1.25 (0.5%) 1.25 (0.5%) 1.25 (0.5%) 1.52 (6.4%) 3.07 (1.3%) 6.542 (27.5%) 164 (0.7%) 254 (1.1%) 1.123 (4.7%) | 0.3% (12%, 0.5%) 0.05 (0.02, 0.07) (;-) 0.01 (0.00, 0.02) (;-) 0.03 (0.01, 0.04) (;-) -0.04 (0.07, -0.01) -(;-) -0.24 (0.21, 0.27) -(;-) 0.1 (0.00, 0.01) 1(;-) 1,-) 1 | 4.137 (28.8%) 2.18 (1.41) 2.20 (1.00, 3.00] 0.00, 4100 1.51 (1.21) 1.00 (1.00, 2.00] 0.00, 3100 0.0 | 219 (1.54) 2.00 (1.00, 3.00) 0.00, 66.00 1.53 (1.20) 1.00 (1.00, 2.00) 0.00, 3.00 0.00 0.00, 3.00 0.00 0.00, 3.00 0.00 0.00 0.00 0.00 0.00 0.00 0.00 | 0.01 (0.04, 0.03) -(-,-) -(-,- |
| HbAIC testsmean (sd)median (lQR)median (lQR)min max Lipid panelsmean (sd)median (lQR)median (lQR)min max Natrivetic peptide testsmean (sd)median (lQR)min maxmedian (lQR)min max | 221(1.44) 2.00 [1.00, 3.00] 0.00, 41.00 1.48 [1.48) 1.00 [1.00, 2.00] 0.00, 1.26 0.0 1.00 [1.00, 2.00] 0.00, 1.26 0.0 0.04 (0.34) 0.00 [1.00, 0.00] 0.00, 2.300 0.12 (0.91) 0.00 [1.00, 0.00] 0.00, 4.00 1.00 0.00, 0.00] 0.00, 4.00 1.00 0.00, 0.00 1.00 0.00, 4.00 1.00 0.00, 0.00 1.00 0.00, 1.00 0.00 0.00, 1.00 0.00 0.00, 1.00 0.00 0.00, 1. | 6,961 (29.3%) 216(1.42) 2.00 [1.00, 3.00] 0.00, 650.0 1.58 (1.18) 1.00 [1.00, 2.00] 0.03, 0.00 0.03, 0.00 0.03, 0.00 0.03, 0.00 0.00 [0.00, 0.00] 0.00 [0.00, 0.00] 0.00 [0.00, 0.00] 0.00 [0.00, 0.00] 0.00 [0.00, 0.00] 0.00, 280.0 0.89 (1.58) 0.00 [0.00, 1.00] 0.03, 34.00 0.93 (1.58) 1.00 [0.00, 2.00] 2.00, 14.00 1.00 [0.00, 2.00] 2.00, 14.00 1.35 [2.05] 0.04 (0.04) 1.35 [2.05] 0.00 [0.00, 0.00] 0.00, 2.700 560 (2.4%) 1.23 [9.2%) 1.25 [9.6%) 1.52 [9.6%] 1.52 [9.6%] | 0.3% (-12%, 0.5%) 0.05 (0.02, 0.07) (-, -) ( | 4.137 (28.8%) 2.18 (1.41) 2.00 (1.00.300] 0.00,410.0 1.51 (1.21) 1.00 (1.00.2.00] 0.00,310.0 0.00,310.0 0.00 (1.00.0.00] 0.00 (1.00.0.0.00] 0.00 (1.00.0.00] 0. | 219 (1.54) 2.09 (1.00, 3.00) 0.00, 66.00 1.53 (1.20) 1.00 (1.00, 2.00] 0.00, 3.00 0.00, | -0.01(-0.04, 0.03) -(-,-) -(-, |
| HbAIC tests | 221(1.44) 2.00 [1.00, 3.00] 0.00, 4100 1.48 [1.48] 1.00 [1.00, 2.00] 0.01, 3.00] 0.01, 3.0 | 6,961 (29.3%) 216(1.42) 2.00 (1.00.3.00) 0.00,66.00 1.58 (1.18) 1.00 (1.00.2.00) 0.00,30.00 0.00,30.00 0.00 (1.00.00) 0.00 (1. | 0.3% (-1.2%, 0.5%) 0.05 (0.02, 0.07) -(-,-) | 4.137 (28.8%) 2.18 (1.41) 2.18 (1.41) 2.00 (1.00, 3.00) 0.00, 41.00 1.51 (1.21) 1.00 (1.00, 2.00) 0.00, 31.00 0.00, 31.00 0.00 (3.00) 0.00 (3.00) 0.00 (0.00, 0.00) 0.00 (0.00, 0.00) 0.00 (0.00, 0.00) 0.00 (0.00, 0.00) 0.00 (0.00, 0.00) 0.00 (0.00, 1.00) 0.00 (0.00, 1.00) 0.00 (1.00, 1.00) 0.00 (1.00 | 219 (1.54) 2.00 (1.00, 3.00) 0.00, 66.00 1.53 (1.20) 1.00 (1.00, 2.00) 0.00, 3.00 0.00 0.00, 3.00 0.00 0.00, 3.00 0.00 0.00 0.00 0.00 0.00 0.00 0.00 | 0.01 (0.04, 0.03) -(-,-) -(-,- |
| HbAIC testsmean (sd)median (lQR)median (lQR)min max Lipid panelsmean (sd)median (lQR)min max Creatinine testsmean (sd)median (lQR)min max Natrivetic peptide testsmean (sd)median (lQR)min maxmedian (lQR)min maxn (sd)min maxn (sd)min maxn (sd)min maxn (sd)min maxn (sd)min maxn (sd)n (sd)n (sd)n (sd)n (sd) | 221(1.44) 2.00 [1.00, 3.00] 0.00, 41.00 1.48 [1.48) 1.00 [1.00, 2.00] 0.00, 1.26 00 1.48 [1.48] 0.00 [1.00, 2.00] 0.00, 1.26 00 0.00, 1.26 00 0.00, 2.30 00 0.00, 2.30 00 0.00, 2.30 00 0.00, 2.30 00 0.00, 2.30 00 0.00, 2.30 00 0.00, 2.30 00 0.00, 0.00 [0.00, 0.00] 0.00, 4.70 00 0.00, 1.00 [0.00, 0.00] 0.00, 1.00 [0.00, 0.00] 0.00, 1.00 [0.00, 1.00] 0.00, 1.00 [0.00, 1.00] 0.00, 1.00 [0.00, 1.00] 0.00, 1.00 [0.00, 1.00] 0.00, 1.00 [0.00, 1.00] 0.00, 1.00 [0.00, 0.00] 0.00, | 6.96I (29.3%) 2.16(1.42) 2.00 [1.00, 3.00] 0.00, 65.00 1.58 (1.18) 1.00 [1.00, 2.00] 0.00, 3.0.00 0.03 (2.5) 0.00 [0.00, 0.00] 0.00 [0.00, 1.00] 0.03 (3.00) 0.03 (3.00) 0.04 (0.01) 0.05 (3.00) 0.05 | 0.3% (12%, 0.5%) 0.05 (0.02, 0.07) -(-,-) - | 4.137 (28.8%) 2.18 (1.41) 2.10 (1.00.300] 0.00, 41.00 1.51 (1.21) 1.00 (1.00.2.00] 0.00, 31.00 0.03 (23) 0.00 (0.00, 0.00] 0.00 (0.00, 0.0 | 219(1.54) 2.09 (1.00, 3.00) 0.00, 66.00 1.53 (1.20) 1.00 (1.00, 2.00] 0.00, 3.00 0.00, 3 | |
| HbAIC tests | 221(1.44) 2.00 [1.00, 3.00] 0.00, 4100 1.48 [1.48] 1.00 [1.00, 2.00] 0.01, 3.00] 0.01, 3.0 | 6,961 (29.3%) 216(1.42) 2.00 (1.00.3.00) 0.00,66.00 1.58 (1.18) 1.00 (1.00.2.00) 0.00,30.00 0.00,30.00 0.00 (1.00.0.00) 0.00 | 0.3% (-1.2%, 0.5%) 0.05 (0.02, 0.07) -(-,-) | 4.137 (28.8%) 2.18 (1.41) 2.18 (1.41) 2.00 (1.00, 3.00) 0.00, 41.00 1.51 (1.21) 1.00 (1.00, 2.00) 0.00, 31.00 0.00, 31.00 0.00 (3.00) 0.00 (3.00) 0.00 (0.00, 0.00) 0.00 (0.00, 0.00) 0.00 (0.00, 0.00) 0.00 (0.00, 0.00) 0.00 (0.00, 0.00) 0.00 (0.00, 1.00) 0.00 (0.00, 1.00) 0.00 (1.00, 1.00) 0.00 (1.00 | 219 (1.54) 2.00 (1.00, 3.00) 0.00, 66.00 1.53 (1.20) 1.00 (1.00, 2.00) 0.00, 3.00 0.00 0.00, 3.00 0.00 0.00, 3.00 0.00 0.00 0.00 0.00 0.00 0.00 0.00 | 0.01 (0.04, 0.03) -(-,-) -(-,- |

Variable\_name

Gender Race

Region

Smoking / Tobacco use Underweight

Normal weight, if BMI is 20.0-24.9 Overweight, if BMI is 25.0 to 29.9

Class 1 (low-risk) obesity, if BMI is 30.0 to 34.9 Class 2 (moderate-risk) obesity, if BMI is 35.0 to 39.9 Class 3 (high-risk) obesity if BMI is equal to or greater than 40 Unspecified obesity

Diabetic retinopathy

Diabetic neuropathy Diabetic nephropathy

Diabetes with other opthalmic complications

Diabetes with peripheral circulatory disorders

Diabetic foot

Erectile dysfuntion

Hypoglycemia

Hyperglycemia/DKA/HONK

Skin infections

Stable angina

Unstable angina

Hypertension

Hypotension

Hyperlipidemia Atrial fibrillation Acute myocardial infarction Old myocardial infarction

Cardiac conduction disorder

Previous cardiac procedure (CABG, PTCA, Stent)

Ischemic stroke PVD diagnosis or surgery

Other cardiac dysrhythmia

Heart failure

Acute heart failure

Microalbuminuria/proteinuria

#### Algorithm sources

If region not available, from State, https://www2.census.gov/geo/pdfs/maps-

data/maps/reference/us\_regdiv.pdf

Investigator review of codes based on:

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015.

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002.

https://pubmed.ncbi.nlm.nih.gov/34953068/.

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9154288/.

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3721171/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/,

https://pubmed.ncbi.nlm.nih.gov/35043165/ Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/,

https://pubmed.ncbi.nlm.nih.gov/35043165/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/ Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/, ICD9 to ICD10 conversion

Investigator review of codes based on:

https://www.ncbi.nlm.nih.gov/books/NBK368403/table/sb203.t5/,

https://www.health.mil/Reference-Center/Publications/2016/03/01/Diabetes-Mellitus,

http://www.icd9data.com/2014/Volume1/240-279/249-259/250/default.htm,

https://www.icd10data.com/ICD10CM/Codes/E00-E89/E08-E13/E11-

Intps://www.icd10data.com/ICD10CM/Codes/N00-N99/N40-N53/N52-,

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4857901/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/,

https://pubmed.ncbi.nlm.nih.gov/35043165/

Investigator review of codes based on:

Hyperglycemia: https://pubmed.ncbi.nlm.nih.gov/34953068/.

https://pubmed.ncbi.nlm.nih.gov/35043165/

DKA: https://pubmed.ncbi.nlm.nih.gov/29773640/. https://pubmed.ncbi.nlm.nih.gov/38262528/

https://dam.assets.ohio.gov/image/upload/medicaid.ohio.gov/Providers/PaymentInnovatio

n/DEF/DKA.pdf

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/ . ICD9

to ICD10 conversion

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/19337843/,

https://pmc.ncbi.nlm.nih.gov/articles/PMC9172873/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/19337843/, https://pmc.ncbi.nlm.nih.gov/articles/PMC9172873/ Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/,

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8929186/

Investigator review of codes based on:

https://pmc.ncbi.nlm.nih.gov/articles/PMC8064679/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/,

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/31933524/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/24682186/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/24682186/ Investigator review of codes based on:

https://stacks.cdc.gov/view/cdc/31381/cdc\_31381\_DS8.pdf,

https://www.health.ny.gov/health\_care/medicaid/redesign/dsrip/vbp\_library/docs/arrblk.pd f, https://www.cdc.gov/dhdsp/maps/atlas/data-sources.html,

https://www.cms.gov/medicare/coding/icd10/downloads/icd10clinicalconceptscardiology1 .pdf, ICD9 to ICD10 conversion

Modified codes based on eligibility criteria, here we implement any care setting, any diagnosis position

Modified codes based on eligibility criteria, here we implement any care setting, any diagnosis position

Investigator review of codes, https://www.icd10data.com/

Investigator review of codes based on:

 $https://stacks.cdc.gov/view/cdc/31381/cdc\_31381\_DS8.pdf,$ 

https://www.health.ny.gov/health\_care/medicaid/redesign/dsrip/vbp\_library/docs/arrblk.pd f, https://www.cdc.gov/dhdsp/maps/atlas/data-sources.html,

https://www.cms.gov/medicare/coding/icd10/downloads/icd10clinicalconceptscardiology1 .pdf, ICD9 to ICD10 conversion

Modified codes based on inclusion criteria, here we implement any care setting, any

diagnosis position Modified codes based on inclusion criteria, here we implement any care setting, any

diagnosis position

Modified codes based on inclusion criteria, here we implement any care setting, any

diagnosis position

Cardiomyopathy Valve disorders Valve replacement TIA Edema Venous thromboembolism/ pulmonary embolsim Pulmonary hypertension Implantable cardioverter defibrillator Hyperkalemia Coronary atherosclerosis Cerebrovascular procedure Insertion of pacemakers / removal of cardiac lead CKD stage 1-2 CKD stage 3-4

Hypertensive nephropathy

Unspecified CKD Acute kidney injury

Urinary tract infections Genital infections

Urolithiasis (kidney or urinary stones)

COPD

Asthma

Obstructive sleep apnea

Serious bacterial infections

Pneumonia

Liver disease

MASH/MASLD

Fractures / Falls

Osteoporosis Osteoarthritis Depression

Dementia

Delirium or psychosis

Anxiety

Sleep disorder

Anemia Influenza

COVID-19

Investigator review of codes based on:

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder mpl2p wn015

Investigator review of codes based on:

https://stacks.cdc.gov/view/cdc/31381/cdc\_31381\_DS8.pdf,

https://pubmed.ncbi.nlm.nih.gov/38440888/

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8751938/,

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015,

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=cder\_mpl2p\_wp009 Modified codes based on eligibility criteria, here we implement any care setting, any diagnosis position

Modified codes based on eligibility criteria, here we implement any care setting, any

diagnosis position

Investigator review of codes based on: https://www.cms.gov/medicare-coveragedatabase/view/article.aspx?articleid=52993&ver=45&

Investigator review of codes based on:

https://www.sciencedirect.com/science/article/pii/S2666572723000251

Investigator review of codes

Modified codes based on eligibility criteria, here we implement any care setting, any diagnosis position

https://pmc.ncbi.nlm.nih.gov/articles/PMC4399109/

Investigator review of codes based on:

https://pmc.ncbi.nlm.nih.gov/articles/PMC10251803/

Investigator review of codes, https://www.icd10data.com/

Modified codes based on eligibility criteria, here we implement any care setting, any diagnosis position

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/

Investigator review of codes based on:

https://pmc.ncbi.nlm.nih.gov/articles/PMC2978782/ Investigator review of codes based on:

https://pmc.ncbi.nlm.nih.gov/articles/PMC5888226/ Investigator review of codes based on:

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8929186/

Investigator review of codes based on:

https://nccd.cdc.gov/ckd/Methods.aspx?Qnum=Q637,

https://www.kidneymedicinejournal.org/cms/10.1016/j.xkme.2022.100414/attachment/5e/second-complex and the complex and the co29ab67-7a7d-4621-9af3-81bd071bbc67/mmc1.pdf,

https://www.icd10data.com/ICD10CM/Codes/I00-I99

Investigator reviewed code based on:

https://pmc.ncbi.nlm.nih.gov/articles/PMC7558992/#app1-antibiotics-09-00536

Investigator reviewed codes based on: https://pubmed.ncbi.nlm.nih.gov/30207042/

Investigator review of codes based on:

https://pmc.ncbi.nlm.nih.gov/articles/PMC7793999/

Investigator review of codes based on:

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10203971/

Investigator review of codes based on:

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10203971/, modified CCW algorithm (any

care setting, any diagnosis position)
Investigator review of codes based on:

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8636332/,

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7927325/

https://pubmed.ncbi.nlm.nih.gov/29921683/, https://pubmed.ncbi.nlm.nih.gov/17346615/,

https://pubmed.ncbi.nlm.nih.gov/23335588/

Investigator review of codes based on:

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10203971/

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002\_

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015, Modified algorightm from\_

https://pubmed.ncbi.nlm.nih.gov/34256144/\_Modified.CCW\_algorithm Investigator review of codes: https://pubmed.ncbi.nlm.nih.gov/32300995/\_

https://pubmed.ncbi.nlm.nih.gov/39316292/

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015,

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

 $packages/browse? at = cder\_mpl2p\_wp009,$ 

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=cder\_mpl2p\_wp010

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8202643/,

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002, CCW Algorithms

Modified CCW algorithm

https://pubmed.ncbi.nlm.nih.gov/35043165/, CCW Algorithms

https://pubmed.ncbi.nlm.nih.gov/35043165/,

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015

https://pubmed.ncbi.nlm.nih.gov/28485014/, https://pubmed.ncbi.nlm.nih.gov/35043165/ ://pubmed.ncbi.nlm.nih.gov/35043165

Investigator review of codes based on https://www.verywellhealth.com/sleeping-disorders-list-anddiagnostic-codes-3014779

Modified codes based on eligibility criteria, here we implement any care setting, any diagnosis position Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/38556924/

https://pubmed.ncbi.nlm.nih.gov/34913208/, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8427377/ Hyperthyroidism and other thyroid gland disorders

Hypothyroidism

Nephrotic syndrome Urinary incontinence

Biliary disease

Pancreatitis

Bowel obstruction Gastroparesis Number of antidiabetic drugs on CED

Concomitant use or initiation of metformin Concomitant use or initiation of insulin

Concomitant use or initiation of sulfonylureas

Concomitant use or initiation of DPP4i

Concomitant use or initiation of SGLT2i

Concomitant use or initiation of other glucose-lowering drugs

Past use of metformin

Past use of insulin

Past use of sulfonylureas

Past use of DPP4i

Past use of SGLT2i

Past use of other glucose-lowering drugs

ACEi / ARB

ARNI

Thiazides

Beta-Blockers

Calcium channel blockers

Digoxin / Digitoxin

Loop diuretics

Other diuretics Intravenous diuretics

Nitrates

Anti-arrhythmics

Statins

PCSK9 inhibitors and other lipid-lowering drugs

Antiplatelet agents

Oral anticoagulants

COPD/Asthma medication

NSAIDs

Oral corticosteroids

Osteoporosis agents (incl. bisphosphonates)

Investigator review of codes based on: https://www.cms.gov/icd10m/version37-fullcodecms/fullcode\_cms/P0244.html

Investigator review of codes based on:

https://pmc.ncbi.nlm.nih.gov/articles/PMC10478599/

 $Investigator\ review\ of\ codes\ based\ on: https://nccd.cdc.gov/ckd/Methods.aspx? Qnum=Q637, and the codes based on the code based on the code based on$ https://www.cms.gov/icd10m/FY2024-nprmversion41.0-fullcode\_cms/P2401.html Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/38527324/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/37796527/, https://pubmed.ncbi.nlm.nih.gov/35851329/,

https://pmc.ncbi.nlm.nih.gov/articles/PMC3985913/,

https://pubmed.ncbi.nlm.nih.gov/38503905/, https://pubmed.ncbi.nlm.nih.gov/35513234/

Investigator review of codes: https://pubmed.ncbi.nlm.nih.gov/36222554/, https://pubmed.ncbi.nlm.nih.gov/30287807/, https://pubmed.ncbi.nlm.nih.gov/22262606/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/36798959/, https://pubmed.ncbi.nlm.nih.gov/28438588/, https://pubmed.ncbi.nlm.nih.gov/31095068/Investigator review of codes: https://pubmed.ncbi.nlm.nih.gov/34624355/

Investigator review of codes

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK518983/ Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK278938/Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK513225/ Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK542331/ Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK576405/ Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK551656/, https://pmc.ncbi.nlm.nih.gov/articles/PMC4882495/, https://www.ncbi.nlm.nih.gov/books/NBK557848/ Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK518983/ Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK278938/

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK513225/Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK542331/ Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK576405/ Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK551656/, https://pmc.ncbi.nlm.nih.gov/articles/PMC4882495/,

https://www.ncbi.nlm.nih.gov/books/NBK557848/ Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/ Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK507904/ Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/ Investigator review of codes, https://www.drugs.com,

https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/lnvestigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/ Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK556025/

https://pubchem.ncbi.nlm.nih.gov/compound/441207 Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/ Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/

Investigator review of codes

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/ Investigator review of codes, https://www.drugs.com,

https://www.ncbi.nlm.nih.gov/books/NBK482322/ (using class I and class II as class 2 is

beta blockers and class 4 is calcium channel blockers)

Investigator review of codes, https://www.drugs.com, https://www.heart.org/en/healthtopics/cholesterol/prevention-and-treatment-of-high-cholesterol-

hyperlipidemia/cholesterol-medications

Investigator review of codes. https://www.drugs.com. https://www.heart.org/en/healthtopics/cholesterol/prevention-and-treatment-of-high-cholesterol-

hyperlipidemia/cholesterol-medications

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK537062/Investigator review of codes, https://www.drugs.com,

https://www.ahajournals.org/doi/full/10.1161/JAHA.120.017559

Investigator review of codes, https://www.copdfoundation.org/Learn-More/l-am-a-Personwith-COPD/Treatments-Medications.aspx, https://getasthmahelp.org/medicationslist.aspx

Investigator review of codes, https://www.drugs.com,

https://www.ncbi.nlm.nih.gov/books/NBK547742/

Investigator review of codes, https://www.drugs.com, https://www.aaaai.org/tools-for-the-

public/drug-guide/oral-corticosteroid-medications Investigator review of codes based on: https://www.drugs.com,

https://www.ncbi.nlm.nih.gov/books/NBK470248/

Opioids

Anti-depressants Antipsychotics

Anxiolytics/hypnotics, benzodiazepines

Medication for dementia Urinary tract infections antibiotics

Laxatives

Number of distinct medications, median (iqr), mean (sd)

Number of office visits median (iqr), mean (sd)

Number of endocrinologist visits, median (iqr), mean (sd)

Number of cardiologist visits, median (iqr), mean (sd)

Number of internal medicine/family medicine visits, median (iqr), mean (sd)

Number of electrocardiograms, median (iqr), mean (sd)

Number of echocardiograms, median (iqr), mean (sd) Pharmacy out-of-pocket cost, median (iqr), mean (sd) Unique brand medications Unique generic medications Ratio of unique brand to generic medications

Colonoscopy/ Sigmoidoscopy

Flu vaccine / Pneumococcal vaccine

Pap smear test

PSA test

Fecal occult blood test Bone mineral density tests

Mammograms

Telemedicine

Number of HbA1c tests, median (iqr), mean (sd) Number of lipid panels, median (iqr), mean (sd) Number of creatinine tests, median (igr), mean (sd) Number of natriuretic peptide tests, median (iqr), mean (sd)

Number of urine tests, median (iqr), mean (sd)

HbA1c Glucose Creatinine

Systolic blood pressure

Heart rate **BMI** eGFR LDL HDL

Total cholesterol Triglycerides

Combined comorbidity score

Investigator review of codes, https://www.drugs.com,

https://pubmed.ncbi.nlm.nih.gov/31643200/#: -: text=They%20can%20also%20be%20information and the state of t

rmally,%2C%20codeine%2C%20oxycodone%2C%20hydrocodone%2C Investigator review of codes, https://www.drugs.com,

https://www.ncbi.nlm.nih.gov/books/NBK538182/

Investigator review of codes, https://www.drugs.com

Investigator review of codes, https://www.drugs.com, https://www.dea.gov/sites/default/files/2020-06/Benzodiazepenes-2020.pdf https://www.ncbi.nlm.nih.gov/books/NBK470159/, https://www.drugs.com Investigator review of codes based on: https://www.drugs.com,

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7462122/,

https://go.drugbank.com/drugs/DB00382

https://pubmed.ncbi.nlm.nih.gov/35790044/ Investigator review of codes, https://www.drugs.com

N/A

https://www.cms.gov/files/document/mm13473-how-use-office-and-outpatient-

evaluation-and-management-visit-complexity-add-code-g2211.pdf,

https://www.cms.gov/files/document/physician-fee-schedule-pfs-payment-

officeoutpatient-evaluation-and-management-em-visits-fact-sheet.pdf
Data dictionary of Optum, Marketscan and https://www.cms.gov/Medicare/ProviderEnrollment-and-Certification/MedicareProviderSupEnroll/downloads/taxonomy.pdf,

https://www.cms.gov/medicare/provider-enrollment-and-

certification/medicareprovidersupenroll/downloads/taxonomycrosswalk.pdf

Data dictionary of Optum, Marketscan and https://www.cms.gov/Medicare/Provider-Enrollment-and-Certification/MedicareProviderSupEnroll/downloads/taxonomy.pdf,

https://www.cms.gov/medicare/provider-enrollment-and-

certification/medicareprovidersupenroll/downloads/taxonomycrosswalk.pdf Data dictionary of Optum, Marketscan and https://www.cms.gov/Medicare/Provider-Enrollment-and-Certification/MedicareProviderSupEnroll/downloads/taxonomy.pdf,

https://www.cms.gov/medicare/provider-enrollment-and-

certification/medicareprovidersupenroll/downloads/taxonomycrosswalk.pdf

https://www.cms.gov/medicare-coverage-database/view/article.aspx?articleld=57326, https://firstcoastbillinggroup.com/ekg-billing-and-reimbursement/,

https://www.aapc.com/codes/coding-newsletters/my-cardiology-coding-alert/cpt-answer-5-common-ecg-coding-questions-175952-article

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8511132/,

https://pubmed.ncbi.nlm.nih.gov/34778785/, https://www.cms.gov/medicare-coverage-

database/view/article.aspx?articleid=56625&ver=27&,

https://www.medicalbillgurus.com/echocardiogram-cpt-code/ N/A

Investigator review of codes, https://www.drugs.com

Investigator review of codes, https://www.drugs.com Investigator review of codes, https://www.drugs.com

packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002

 $https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=refs%2Fheads%2Fcder_sir_wp002, https://www.cms.gov/medicare-coverage-database/view/article.aspx?articleld=54767&DocID=A54767, https://www.cms.gov/medicare-coverage-database/view/article.aspx.gov/medicare-coverage-database/vi$ 

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002, https://www.cms.gov/medicare-

coverage-database/view/article.aspx?articleId=54767&DocID=A54767

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002, http://www.icd9data.com/2012/Volume1/V01-V91/V70-V82/V72/default.htm,

http://www.icd9data.com/2012/Volume1/V01-V91/V70-V82/V76/default.htm

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-

packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002

Investigator review of codes

N/A

Investigator review of codes based on:

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002, https://www.cms.gov/medicare-

coverage-database/view/article.aspx?articleid=56448&ver=16&bc=0,

http://www.icd9data.com/2012/Volume1/V01-V91/V70-V82/V76/default.htm

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/33151319/,

https://www.cms.gov/newsroom/fact-sheets/medicare-telemedicine-health-care-provider-factsheet, https://www.aafp.org/family-physician/practice-and-career/getting-paid/coding/coding-

telehealth-audio-virtual-digital-visits.html https://pubmed.ncbi.nlm.nih.gov/34953068/

https://pubmed.ncbi.nlm.nih.gov/34953068/

https://pubmed.ncbi.nlm.nih.gov/34953068/

Investigator review of codes Investigator review of codes

N/A

N/A

N/A

N/A N/A

N/A

N/A

N/A

N/A

A combined comorbidity score predicted mortality in elderly patients better than existing

scores, https://pubmed.ncbi.nlm.nih.gov/21208778/

Frailty score Fraitty score
Number of any hospitalization, median (iqr), mean (sd)
Any hospitalization within prior 90 days; n (%)
Any hospitalization within prior 91-365 days; n (%)
0, 1, >1 hospitalizations (any) Hospitalization for heart failure; n (%)

Number of emergency department visit median (iqr), mean (sd) Calendar year

Measuring Frailty in Medicare Data: Development and Validation of a Claims-Based Frailty Index, https://pubmed.ncbi.nlm.nih.gov/29244057/N/A

N/A N/A N/A N/A

Different in all 3 databases and measure already created in all 3 as well; ED visit (Medicare): Revenue center codes: 0450, 0451, 0452, 0456, 0459, 0981; Place

ED visit (Wetchae): Nevertide Center Codes. 0430, 0431, 0432, 0430, 0433, 0431, 11ace of service: 23

ED visit (Optum): Place of service: 23

ED visit (Marketscan): Service sub-category codes: 10120, 10220, 10320, 10420, 10520, 12220, 20120, 20220, 21120, 21220, 22120, 22320, 30120, 30220, 30320, 30420, 30520, 30620, 31120, 31220, 31320, 31420, 31520, 31620; Place of service: 23

# TIRZSEMA-CVOT- TIRZSEMA

# **Appendices**

| 1 | Target Trial Framework, Operational Definitions and Data Fitness Assessment |
|---|---|
| 2 | Codealgorithms |
| 2a | Exposure |
| 2b | Inclusion |
| 2c | Exclusion |
| 2d | Outcome |
| 3 | Flowchart for cohort assembly |
| 4 | 1st feasibility assessment |
| 5 | 2nd feasibility assessment |
| 6 | Balance Assessment - PS Distribution and C-Statistic |
| 7 | Balance Assessment - Table 1 |
| 8 | Covariate - Algorithm Sources |

| | TIRZSEMA | OPTUM | MARKETSCAN | Notes/Questions |
|---|---|---|---|---|
| | International, double-blind, randomized, active-controlled trial to treatment A vs B $$ | Non-randomized initiation of treatment Tirzepatide vs Semaglutide (first eligible entry to study population) | Non-randomized initiation of treatment Tirzepatide vs Semaglutide (first eligible entry to study population) | G |
| index date) | trial to treatment A VS B | Code type: RX | Code type: RX | G |
| | | Care setting: N/A | Care setting: N/A | |
| | | Diagnosis position: N/A Washout window: [-183,-1] | Diagnosis position: N/A Washout window: [-183, -1] | |
| | | Incident with respect to: Tirzepatide in any formulation or dose | Incident with respect to: Tirzepatide in any formulation or dose | |
| | Tirzepatide (subcutaneously | Assessment window: N/A Source of algorithm: N/A | Assessment window: N/A Source of algorithm: N/A | |
| | once per week) | Measurement characteristics: N/A | Measurement characteristics: N/A | М |
| | | Code type: RX Care setting: N/A | Code type: RX Care setting: N/A | |
| | | Diagnosis position: N/A | Diagnosis position: N/A | |
| | | Washout window: [-183, -1] Incident with respect to: Dulaglutide in any formulation or dose | Washout window: [-183,-1] Incident with respect to: Dulaglutide in any formulation or dose | |
| | | Assessment window: N/A | Assessment window: N/A | |
| Comparator | Semaglutide (subcutaneously once per week) | Source of algorithm: N/A Measurement characteristics: N/A | Source of algorithm: N/A Measurement characteristics: N/A | Po |
| • | | Code type: DX, PX | Code type: DX, PX | |
| | | Care setting: Inpatient for stroke/MI, any for death Diagnosis position: Primary for Stroke, Any for MI | Care setting: Inpatient for stroke/MI, any for death Diagnosis position: Primary | |
| | | Washout window: Source of algorithm: Measurement characteristics: Death includes information | Washout window: Source of algorithm: Measurement characteristics: Death includes information | |
| | | from the inpatient discharged dead status, social security death master file, and | from the inpatient discharged dead status, social security death master file, and | Pe |
| Primary outcome to be emulated | MACE, defined as CV death, MI, or stroke | deaths scraped from obituaries or other sources. Code type: DX. PX | deaths scraped from obituaries or other sources. Code type: DX. PX | in |
| | | Care setting: Inpatient for stroke/MI/ heart failure, any for death, outpatient for i.v. | | |
| | | diuretics Diagnosis position: Primary for stroke/ heart failure, any for MI | diuretics Diagnosis position: Primary for stroke/ heart failure, any for MI | |
| | | Washout window: | Washout window: | |
| | | Source of algorithm: PROMISE Team, Validation studies, (Investigator reviewed codes) | Source of algorithm: PROMISE Team, Validation studies, (Investigator reviewed codes) | |
| | | Measurement characteristics: Death includes information from the inpatient | Measurement characteristics: Death includes information from the inpatient | |
| | | discharged dead status, social security death master file, and deaths scraped from<br>obituaries or other sources. | discharged dead status, social security death master file, and deaths scraped from obituaries or other sources. | |
| | | PPV for ischemic stroke using ICD9 codes was 88% and 95% [https://pubmed.ncbi.nlm.nih.gov/12364739/ and | PPV for ischemic stroke using ICD9 codes was 88% and 95% [https://pubmed.ncbi.nlm.nih.gov/12364739/ and | |
| | - Individual components of the primary endpoint, i.e., all- | https://pubmed.ncbi.nlm.nih.gov/20140892/] | https://pubmed.ncbi.nlm.nih.gov/20140892/] | |
| | cause mortality, myocardial infarction, or stroke. - Composite of all-cause mortality, hospitalization for | Both of the above ICD9 codes were mapped to ICD10, but no validation study was performed. | Both of the above ICD9 codes were mapped to ICD10, but no validation study was performed. | |
| | heart failure, or urgent heart failure visits requiring | PPV for HHF diagnosis using ICD-10 codes was 98% in a national Medicare | PPV for HHF diagnosis using ICD-10 codes was 98% in a national Medicare | |
| | intravenous diuretics. Randomization date | sample. One day after initiation of treatment with tirzepatide or dulaglutide | sample. One day after initiation of treatment with tirzepatide or dulaglutide | |
| rollow up start | Nandomization date | Earliest of: Outcome, end of observation in data, end of study period (365 days), | Earliest of: Outcome, end of observation in data, end of study period (365 days), | |
| Follow up end | 1 year | discontinuation of study drug (45 days grace window and risk-window), switch to other GLP-1-RA, nursing home admission | discontinuation of study drug (45 days grace window and risk-window), switch to other GLP-1-RA, nursing home admission | |
| | | | | Algorithm detail: Adherence in clinical practice databases is |
| | | | | expected to be much worse than in the trial, therefore the on-<br>treatment analysis at 1 year follow-up will be the primary |
| | Intention-to-treat effect Cox proportional hazards model | On-treatment effect Cox proportional hazards regression model | On-treatment effect Cox proportional hazards regression model | analysis. |
| Inclusion criteria | COX proportional nazards model | | | |
| | | Applied before/after selection of index date: Before Assessment window: [0, 0] | Applied before/after selection of index date: Before Assessment window: [0, 0] | |
| | | Code type: N/A | Code type: N/A | |
| | | Care setting: N/A Diagnosis position: N/A | Care setting: N/A Diagnosis position: N/A | |
| | | Source of algorithm: N/A | Source of algorithm: N/A | |
| 1 | Men and women aged 18 years or older | Measurement characteristics: N/A Applied before/after selection of index date: Before | Measurement characteristics: N/A Applied before/after selection of index date: Before | |
| | | Assessment window: [-365,0] | Assessment window: [-365, 0] | |
| | | Code type: DX Care setting: Any | Code type: DX Care setting: Any | |
| | | Diagnosis position: Any Source of algorithm: PROMISE team | Diagnosis position: Any Source of algorithm: PROMISE team | |
| 2 | Type 2 diabetes mellitus | Measurement characteristics: N/A | Measurement characteristics: N/A | |
| | | Applied before/after selection of index date: Before Assessment window: [-730, 0] | Applied before/after selection of index date: Before Assessment window: [-730, 0] | |
| | | Code type: DX, LOINC | Code type: DX, LOINC | |
| | | Care setting: Any Diagnosis position: Any | Care setting: Any Diagnosis position: Any | |
| | | Source of algorithm: Validation of obesity-related diagnosis codes in claims data; Validation of body mass index (BMI)-related ICD-9-CM and ICD-10-CM | Source of algorithm: Validation of obesity-related diagnosis codes in claims | |
| | | administrative diagnosis codes recorded in US claims data | data: Validation of body mass index (BMI)-related ICD-9-CM and ICD-10-CM administrative diagnosis codes recorded in US claims data | Algorithm detail: If BMI measurement via LOINC code is |
| | BMI ≥ 25kg/m2 | Measurement characteristics: N/A | Measurement characteristics: N/A | below 10 or above 100 then measurent is set to missing. |
| | Low, moderate, or high cardiovascular risk, definded a<br>History of a cardiovascular event | | | |
| | | Applied before/after selection of index date: Before Assessment window: [all available data, 0] | Applied before/after selection of index date: Before Assessment window: [all available data, 0] | |
| | | Code type: DX | Code type: DX | |
| | | Care setting: Any Diagnosis position: Any | Care setting: Any Diagnosis position: Any | |
| | Documented history of myocardial infarction or unstable | Source of algorithm: N/A | Source of algorithm: N/A | |
| 4.1.1 | angina | Measurement characteristics: N/A | Measurement characteristics: N/A | |

**Color coding** 

Good proxy definition

Moderate proxy definition

Poorly measured in database

Poorly measured in database and not

| | | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before |
|---|---|---|---|
| | | Assessment window: [all available data, 0] | Assessment window: [all available data, 0] |
| | | Code type: DX | Code type: DX |
| | | Care setting: Any Diagnosis position: Any | Caresetting: Any Diagnosis position: Any |
| | | Source of algorithm: N/A | Source of algorithm: N/A |
| 4.1.2 | History of ischemic stroke or TIA | Measurement characteristics: N/A | Measurement characteristics: N/A |
| | , | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before |
| | | Assessment window: [all available data, 0] | Assessment window: [all available data, 0] |
| | | Code type: DX | Code type: DX |
| | | Care setting: Any | Care setting: Any |
| | | Diagnosis position: Any | Diagnosis position: Any |
| | | Source of algorithm: DUPLICATE team, investigator reviewed codes | Source of algorithm: DUPLICATE team, investigator reviewed codes |
| 4.1.3 | History of heart failure | Measurement characteristics: N/A | Measurement characteristics: N/A |
| | | Applied before/after selection of index date: Before Assessment window: [all available data, 0] | Applied before/after selection of index date: Before Assessment window: [all available data, 0] |
| | | Code type: DX | Code type: DX |
| | | Care setting: Any | Care setting: Any |
| | | Diagnosis position: Any | Diagnosis position: Any |
| | History of surgical or percutaneous coronary | Source of algorithm: PROMISE team | Source of algorithm: PROMISE team |
| 4.1.4 | revascularization procedure | Measurement characteristics: N/A | Measurement characteristics: N/A |
| | | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before |
| | | Assessment window: [all available data, 0] | Assessment window: [all available data, 0] |
| | | Code type: DX, PX Care setting: Any | Code type: DX, PX<br>Care setting: Any |
| | | Diagnosis position: Any | Diagnosis position: Any |
| | | Source of algorithm: N/A | Source of algorithm: N/A |
| 4.1.5 | History of carotid stenting or surgical revascularization | Measurement characteristics: N/A | Measurement characteristics: N/A |
| | | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before |
| | | Assessment window: [all available data, 0] | Assessment window: [all available data, 0] |
| | | Code type: DX, PX | Code type: DX, PX |
| | | Care setting: Any | Caresetting: Any |
| | Illestern of a relational constraint and the fet of the second | Diagnosis position: Any | Diagnosis position: Any |
| 416 | History of peripheral vascular procedure (stenting or<br>surgical revascularization) | Source of algorithm: N/A Measurement characteristics: N/A | Source of algorithm: N/A Measurement characteristics: N/A |
| 4.1.0 | surgicarrevascularizationij | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before |
| | | Assessment window: [all available data, 0] | Assessment window: [all available data, 0] |
| | | Code type: RX | Code type: RX |
| | | Care setting: N/A | Care setting: N/A |
| | | Diagnosis position: N/A | Diagnosis position: N/A |
| | | Source of algorithm: Primary agents as defined by ACC/AHA guidelines for high | Source of algorithm: Primary agents as defined by ACC/AHA guidelines for high |
| 4.0 | 0 6 1 11 1 1 | blood pressure | blood pressure |
| 4.2 | Current use of ≥1 antihypertensive drug | Measurement characteristics: N/A Applied before/after selection of index date: Before | Measurement characteristics: N/A Applied before/after selection of index date: Before |
| | | Assessment window: [all available data, 0] | Assessment window: [all available data, 0] |
| | | Code type: RX | |
| | | Codetype: RX Care setting: N/A | Code type: RX |
| | | Care setting: N/A Diagnosis position: N/A | |
| | | Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by | Code type: RX Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by |
| | | Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA guidelines on management of blood cholesterol. | Code type: RX Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA audicelines on management of blood cholesterol |
| | Current use of ≥1 lipid-lowering drug | Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by | Code type: RX Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by |
| | Current use of ≥1 lipid-lowering drug<br>History of atherosclerotic cardiovascular disease | Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suidelines on management of blood cholesterol Measurement characteristics: N/A | Code type: RX Care setting: N/A Diagnosis position: N/A Sugnosis position: N/A Sugnosis position: N/A Succidant audelines on management of blood cholesterol Measurement characteristics: N/A |
| | | Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suidelines on management of blood cholesterol Measurement characteristics: N/A Applied before/after selection of index date: Before | Code type: RX Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA guidelines on management of blood cholesterol Measurement characteristics: N/A Applied before/after selection of index date: Before |
| | | Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suidelines on management of blood cholesterol Measurement characteristics: N/A | Code type: RX Care setting: N/A Diagnosis position: N/A Sugnosis position: N/A Sugnosis position: N/A Succidant audelines on management of blood cholesterol Measurement characteristics: N/A |
| | | Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suddelines on management of blood cholesterol Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any | Code type: RX Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA studelines on manuscement of blood cholesterol Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any |
| | | Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suddelines on management of blood cholesterol. Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: D/X Care setting: Any Diagnosis position: Any | Code type: RX Care setting: N/A Diagnosis position: N/A Sugnosis position: N/A Sugnosis position: N/A Sugnosis position: N/A Succi Alfa Agudelines on management of blood cholesterol Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any |
| 4.4 | History of atherosclerotic cardiovascular disease | Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suddelines on management of blood cholesterol. Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Codetype: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A | Code type: RX Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suddelines on management of blood cholesterol Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A |
| 4.4 | | Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA exidelines on management of blood cholesterol Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: D/X Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A | Code type: RX Diagnosis position: N/A Diagnosis position: N/A Sugnosis position: N/A Succept algorithm: Common lipid-lowering medications as defined by Succept algorithm: One of algorithm: One of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A |
| 4.4 | History of atherosclerotic cardiovascular disease | Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suidelines sommanasement of blood cholesterol Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before | Code type: RX Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suddelines on management of blood cholesterol Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Measurement characteristics: N/A |
| 4.4 | History of atherosclerotic cardiovascular disease | Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suddelines on management of blood cholesterol Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] | Code type: RX Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suitelines on management of blood cholesterol Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Core setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] |
| 4.4 | History of atherosclerotic cardiovascular disease | Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suddelines on management of blood cholesterol. Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Care setting: Any | Code type: RX Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA-autelines on manuscement of blood cholesterol Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Measurement window: [all available data, 0] Code type: DX |
| 4.4 | History of atherosclerotic cardiovascular disease | Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suidclines on manuscement of blood cholesterol. Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Surces DX Care setting: Any Diagnosis position: Any | Code type: RX Diagnosis position: R/A Diagnosis position: R/A Diagnosis position: R/A Diagnosis position: R/A Succi Alfa Agudelines on management of blood cholesterol Measurement characteristics: R/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Care setting: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any |
| 4.4.1 | History of atherosclerotic cardiovascular disease Documented history of coronary artery disease | Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suidelines on management of blood cholesterol. Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: D/X Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: D/X Care setting: Any Diagnosis position: Any Source of algorithm: N/A | Code type: RX Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suitelines on manuscement of blood cholesterol Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Manuscharacteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A |
| 4.4.1 | History of atherosclerotic cardiovascular disease | Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suddelines on mensurement of blood cholesterol. Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Measurement characteristics: N/A Measurement characteristics: N/A Measurement characteristics: N/A Measurement characteristics: N/A | Code type: RX Diagnosis position: N/A Diagnosis position: N/A Diagnosis position: N/A Diagnosis position: N/A Succi Alfa Rudelines on management of blood cholesterol Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Source of algorithm: N/A Measurement characteristics: N/A Measurement characteristics: N/A Measurement characteristics: N/A |
| 4.4.1 | History of atherosclerotic cardiovascular disease Documented history of coronary artery disease | Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suidelines on management of blood cholesterol Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before | Code type: RX Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA statellines on management of blood cholesterol Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: n/A Applied before/after selection of index date: Before |
| 4.4.1 | History of atherosclerotic cardiovascular disease Documented history of coronary artery disease | Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA eudelines on management of blood cholesterol. Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment tharacteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] | Code type: RX Diagnosis position: N/A Diagnosis position: N/A Diagnosis position: N/A Succo falgorithm: Common lipid-lowering medications as defined by Succo falgorithm: Common lipid-lowering medications as defined by Succo falgorithm: Common lipid-lowering medications as defined by Succo falgorithm: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] |
| 4.4.1 | History of atherosclerotic cardiovascular disease Documented history of coronary artery disease | Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suitediness or manascerner of blood cholesterol Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: Office of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX | Code type: RX Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suddelines on management of blood cholesterol Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX X |
| 4.4.1 | History of atherosclerotic cardiovascular disease Documented history of coronary artery disease | Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA eudelines on management of blood cholesterol. Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Care setting: Any Care setting: Any | Code type: RX Diagnosis position: N/A Diagnosis position: N/A Diagnosis position: N/A Succo falgorithm: Common lipid-lowering medications as defined by SCCC/AHA suitelines on management of blood cholesterol Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any |
| 4.4.1<br>4.4.2 | History of atherosclerotic cardiovascular disease Documented history of coronary artery disease Documented history of carotid artery disease | Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA exidelines on management of blood cholesterol. Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any | Code type: RX Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA-autidines on management of blood cholesterol Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Core type: DX Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Code type: DX Core setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Core of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Core of selecting: Any Diagnosis position: Any Source of algorithm: N/A Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: N/A |
| 4.4.1<br>4.4.2<br>4.4.3 | History of atherosclerotic cardiovascular disease Documented history of coronary artery disease | Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suitediness on manuscement of blood cholesterol. Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Juganosis position: Any | Code type: RX Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suddelines on management of blood cholesterol Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Measurement window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Measur |
| 4.4.1<br>4.4.2 | History of atherosclerotic cardiovascular disease Documented history of coronary artery disease Documented history of carotid artery disease | Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA evidelines on management of blood cholesterol. Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Measurement characteristics: N/A Measurement characteristics: N/A Measurement characteristics: N/A Measurement characteristics: N/A Source of algorithm: N/A Measurement characteristics: N/A Source of algorithm: N/A Source of algorithm: N/A Source of algorithm: N/A Diagnosis position: Any Source of algorithm: N/A Source of algorithm: N/A Measurement characteristics: N/A | Code type: RX Diagnosis position: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suddelines on manuscement of blood cholesterol Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Measurement characteristics: N/A Measurement characteristics: N/A Measurement characteristics: N/A Measurement window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Care setting: Any Diagnosis position: Any Source of algorithm: N/A Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Measurement characteristics: N/A Measurement characteristics: N/A |
| 4.4.1<br>4.4.2<br>4.4.3 | History of atherosclerotic cardiovascular disease Documented history of coronary artery disease Documented history of carotid artery disease | Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suddelines on management of blood cholesterol. Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: D/X Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: D/X Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: D/X Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement window: [all available data, 0] Code type: D/X Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Measurement characteristics: N/A Applied before/after selection of index date: Before | Code type:RX Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suddelines on management of blood cholesterol Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before |
| 4.4.1<br>4.4.2<br>4.4.3 | History of atherosclerotic cardiovascular disease Documented history of coronary artery disease Documented history of carotid artery disease | Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suitediness on manascented foliood cholesterol Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: D/X Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: D/X Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: D/X Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] | Code type: RX Diagnosis position: N/A Diagnosis position: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA standardines on management of blood cholesterol Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] |
| 4.4.1<br>4.4.2<br>4.4.3 | History of atherosclerotic cardiovascular disease Documented history of coronary artery disease Documented history of carotid artery disease | Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA eudelines on management of blood cholesterol. Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A | Code type: RX Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suidelines on management of blood cholesterol Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Core setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX |
| 4.4.1<br>4.4.2<br>4.4.3 | History of atherosclerotic cardiovascular disease Documented history of coronary artery disease Documented history of carotid artery disease | Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA eudelines on management of blood cholesterol. Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of position: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any | Code type: RX Diagnosis position: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suitedines on management of blood cholesterol Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any |
| 4.4.1 4.4.2 4.4.3 Exclusion criteria | History of atherosclerotic cardiovascular disease Documented history of coronary artery disease Documented history of carotid artery disease Documented history of peripheral artery disease | Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suitediness on manascement of blood cholesterol. Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: D/X Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: D/X Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: D/X Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: D/X Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: D/X Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team | Code type:RX Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suddelines on management of blood cholesterol Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Core setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Measurement characteristics: N/A Measurement daracteristics: N/A Measurement daracteristics: N/A Measurement characteristics: N/A Measurement char |
| 4.4.1 4.4.2 4.4.3 Exclusion criteria | History of atherosclerotic cardiovascular disease Documented history of coronary artery disease Documented history of carotid artery disease | Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA eudelines on management of blood cholesterol. Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A | Code type: RX Diagnosis position: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA-autidines on manuscement of blood cholesterol Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A |
| 4.4.1 4.4.2 4.4.3 Exclusion criteria | History of atherosclerotic cardiovascular disease Documented history of coronary artery disease Documented history of carotid artery disease Documented history of peripheral artery disease | Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suidelines on manascement of blood cholesterol. Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A | Code type: RX Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suddelines on management of blood cholesterol Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Core setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PKOMISE team Measurement characteristics: N/A |
| 4.4.1 4.4.2 4.4.3 Exclusion criteria | History of atherosclerotic cardiovascular disease Documented history of coronary artery disease Documented history of carotid artery disease Documented history of peripheral artery disease | Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA evadelines on management of blood cholesterol. Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Source of algorithm: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Source of algorithm: W/A Applied before/after selection of index date: Before Assessment window: [-365, 0] | Code type: RX Diagnosis position: VIA Diagnosis position: VIA Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA-autidines on management of blood cholesterol Measurement characteristics: VIA Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] |
| 4.4.1 4.4.2 4.4.3 Exclusion criteria | History of atherosclerotic cardiovascular disease Documented history of coronary artery disease Documented history of carotid artery disease Documented history of peripheral artery disease | Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suddelines on mensurement of blood cholesterol. Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Mepside before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Mepside before/after selection of index date: Before Assessment window: [-310, 0] Code type: DX Code type | Code type: RX Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suitelines on management of blood cholesterol Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Measurement characteristics: N/A Measurement characteristics: N/A Measurement characteristics: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX |
| 4.4.1 4.4.2 4.4.3 Exclusion criteria | History of atherosclerotic cardiovascular disease Documented history of coronary artery disease Documented history of carotid artery disease Documented history of peripheral artery disease | Care setting: Any Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA evidelines on management of blood cholesterol. Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any | Code type: RX Diagnosis position: VIA Diagnosis position: VIA Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suitelines on manuscement of blood cholesterol Measurement characteristics: VIA Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: VIA Measurement characteristics: NIA Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: NIA Measurement characteristics: NIA Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: NIA Measurement characteristics: NIA Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: NIA Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: NIA Applied before/after selection of index date: Before Assessment window: [-305, 0] Code type: DX Care setting: Any |
| 4.4.1 4.4.2 4.4.3 Exclusion criteria | History of atherosclerotic cardiovascular disease Documented history of coronary artery disease Documented history of carotid artery disease Documented history of peripheral artery disease History of T1DM or secondary diabetes | Care setting: N/A Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suddelines on mensurement of blood cholesterol. Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Measurement characteristics: N/ | Code type: RX Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suddelines on management of blood cholesterol Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any |
| 4.4.1 4.4.2 4.4.3 Exclusion criteria | History of atherosclerotic cardiovascular disease Documented history of coronary artery disease Documented history of carotid artery disease Documented history of peripheral artery disease | Care setting: Any Diagnosis position: N/A Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA evidelines on management of blood cholesterol. Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any | Code type: RX Diagnosis position: VIA Diagnosis position: VIA Source of algorithm: Common lipid-lowering medications as defined by ACC/AHA suitelines on manuscement of blood cholesterol Measurement characteristics: VIA Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: VIA Measurement characteristics: NIA Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: NIA Measurement characteristics: NIA Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: NIA Measurement characteristics: NIA Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: NIA Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: NIA Applied before/after selection of index date: Before Assessment window: [-305, 0] Code type: DX Care setting: Any |

| | | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | |
|---|---|---|---|---|
| | | Assessment window: [-365, 0] | Assessment window: [-365,0] | |
| | | Code type: DX, PX | Code type: DX, PX | |
| | | Care setting: Any | Care setting: Anv | |
| | | Diagnosis position: Any | Diagnosis position: Any | Algorithm detail: Proxied by ICD-10-CM codes for chronic |
| | | Source of algorithm: PROMISE team | Source of algorithm: PROMISE team | kidney disease stage 5 OR end-stage renal disease OR ICD- |
| 7 | End-stage renal disease or dialysis | Measurement characteristics: N/A | Measurement characteristics: N/A | 10-CM procedure codes for dialysis. |
| | | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | |
| | | Assessment window: [-365, 0] | Assessment window: [-365, 0] | |
| | | Code type: PX | Code type: PX | |
| | | Care setting: Any | Care setting: Any | |
| | | Diagnosis position: Any | Diagnosis position: Any | Algorithm detail: Will be proxied by a history of treatment |
| | History of treatment for diabetic retinopathy and/or | Source of algorithm: PROMISE team | Source of algorithm: PROMISE team | (e.g. codes for intravitreal injection of anti-VEGFi OR |
| 8 | macular edema | Measurement characteristics: N/A | Measurement characteristics: N/A | photocoagulation.) |
| | | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | |
| | | Assessment window: [all available data, 0] | Assessment window: [all available data, 0] | |
| | | Code type: DX | Code type: DX | |
| | | Care setting: Any | Care setting: Any | |
| | | Diagnosis position: Any | Diagnosis position: Any | |
| | | Source of algorithm: PROMISE team | Source of algorithm: PROMISE team | |
| 9 | History of any malignancy | Measurement characteristics: N/A | Measurement characteristics: N/A | |
| | | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | |
| | | Assessment window: [-7, 0] | Assessment window: [-7, 0] | |
| | | Code type: DX, PX | Code type: DX, PX | |
| | | Care setting: Inpatient/ED for MI, Stroke, TIA, inpatient for procedures | Care setting: Inpatient/ED for MI, Stroke, TIA, inpatient for procedures | |
| | | Diagnosis position: Any | Diagnosis position: Any | |
| | | Source of algorithm: PROMISE team, Investigator reviewed codes | Source of algorithm: PROMISE team, Investigator reviewed codes | |
| 10 | Cardiovascular event or intervention in the past 7 days | Measurement characteristics: N/A | Measurement characteristics: N/A | |
| | | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | |
| | | Assessment window: [-365, 0] | Assessment window: [-365, 0] | |
| | | Code type: DX | Code type: DX | |
| | | Care setting: Any | Care setting: Any | |
| | | Diagnosis position: Any | Diagnosis position: Any | |
| | Wassessels and a second a second and a second a second and a second a | Source of algorithm: Pregnancy team Measurement characteristics: N/A | Source of algorithm: Pregnancy team Measurement characteristics: N/A | Algorithm detail: Proxied by ICD-10-CM codes indicative of |
| 11 | Women who are pregnant or breastfeeding | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | pregnancy at baseline. |
| | | Assessment window: [-183, 0] | Assessment window: [-183,0] | |
| | | Code type: RX | Code type: RX | |
| | | Care setting: N/A | Care setting: N/A | |
| | | Diagnosis position: N/A | Diagnosis position: N/A | |
| | | Source of algorithm: N/A | Source of algorithm: N/A | |
| 12 | GLP-1-RA treatment within past 6 months | Measurement characteristics: n/a | Measurement characteristics: n/a | |
| | der 2 tota danient wantpast officials | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | |
| | | Assessment window: [-365,0] | Assessment window: [-365, 0] | |
| | | Code type: PX | Code type: PX | |
| | | Care setting: Any | Care setting: Anv | |
| | | Diagnosis position: Any | Diagnosis position: Any | |
| | | Source of algorithm: PROMISE team | Source of algorithm: PROMISE team | |
| 13 | Bariatric surgery within the past 12 months | Measurement characteristics: N/A | Measurement characteristics: N/A | |


| TIA |
|-----|


| REOPERATION, CORONARY ARTERY BYPASS PROCEDURE OR VALVE | |
|---|---|
| History of surgical or PROCEDURE, MORE THAN 1 MONTH AFTER ORIGINAL OPERATION | |
| percutaneous coronary (LIST SEPARATELY IN ADDITION TO CODE FOR PRIMARY 4.1.4 revascularization procedure 33530 PX PROCEDURE) ICD-1 | 0-PCS |
| History of surgical or | 0-PC3 |
| percutaneous coronary CORONARY ARTERY BYPASS, USING ARTERIAL GRAFT(S); SINGLE | |
| | 0-PCS |
| History of surgical or CORONARY ARTERY BYPASS, USING ARTERIAL GRAFT(S); 2 | |
| | 0-PCS |
| History of surgical or | |
| percutaneous coronary CORONARY ARTERY BYPASS, USING ARTERIAL GRAFT(S); 3 | 0 000 |
| <b>4.1.4</b> revascularization procedure 33535 PX CORONARY ARTERIAL GRAFTS ICD-1 History of surgical or | 0-PCS |
| percutaneous coronary CORONARY ARTERY BYPASS, USING ARTERIAL GRAFT(S); 4 OR MORE | |
| | 0-PCS |
| History of surgical or | |
| percutaneous coronary 4.1.4 revascularization procedure 33545 PX REPAIR OF POSTINFARCTION VENTRICULAR SEPTAL DEFECT, WITH OR WITHOUT MYOCARDIAL RESECTION ICD-1 | 0-PCS |
| CORONARY ENDARTERECTOMY, OPEN, ANY METHOD, OF LEFT | 0-FC3 |
| ANTERIOR DESCENDING, CIRCUMFLEX, OR RIGHT CORONARY | |
| History of surgical or ARTERY PERFORMED IN CONJUNCTION WITH CORONARY ARTERY | |
| percutaneous coronary BYPASS GRAFT PROCEDURE, EACH VESSEL (LIST SEPARATELY IN 4.1.4 revascularization procedure 33572 PX ADDITION TO PRIMARY PROCEDURE) ICD-1 | 0-PCS |
| History of surgical or | 0-663 |
| percutaneous coronary PERCUTANEOUS TRANSLUMINAL CORONARY ANGIOPLASTY; SINGLE | |
| | 0-PCS |
| History of surgical or PERCUTANEOUS TRANSLUMINAL CORONARY ANGIOPLASTY; EACH percutaneous coronary ADDITIONAL BRANCH OF A MAJOR CORONARY ARTERY (LIST | |
| | 0-PCS |
| History of surgical or PERCUTANEOUS TRANSLUMINAL CORONARY ATHERECTOMY, WITH | |
| percutaneous coronary CORONARY ANGIOPLASTY WHEN PERFORMED; SINGLE MAJOR | 0 000 |
| <b>4.1.4</b> revascularization procedure 92924 PX CORONARY ARTERY OR BRANCH ICD-1 PERCUTANEOUS TRANSLUMINAL CORONARY ATHERECTOMY, WITH | 0-PCS |
| History of surgical or CORONARY ANGIOPLASTY WHEN PERFORMED; EACH ADDITIONAL | |
| percutaneous coronary BRANCH OF A MAJOR CORONARY ARTERY (LIST SEPARATELY IN | |
| <b>4.1.4</b> revascularization procedure 92925 PX ADDITION TO CODE FOR PRIMARY PROCEDURE) ICD-1 | 0-PCS |
| History of surgical or PERCUTANEOUS TRANSCATHETER PLACEMENT OF | |
| percutaneous coronary INTRACORONARY STENT(S), WITH CORONARY ANGIOPLASTY WHEN | |
| | 0-PCS |
| PERCUTANEOUS TRANSCATHETER PLACEMENT OF INTRACORONARY STENT(S), WITH CORONARY ANGIOPLASTY WHEN | |
| History of surgical or PERFORMED; EACH ADDITIONAL BRANCH OF A MAJOR CORONARY | |
| percutaneous coronary ARTERY (LIST SEPARATELY IN ADDITION TO CODE FOR PRIMARY | |
| <b>4.1.4</b> revascularization procedure 92929 PX PROCEDURE) ICD-1 | 0-PCS |
| History of surgical or PERCUTANEOUS TRANSLUMINAL CORONARY ATHERECTOMY, WITH | |
| percutaneous coronary INTRACORONARY STENT, WITH CORONARY ANGIOPLASTY WHEN | |
| | 0-PCS |
| PERCUTANEOUS TRANSLUMINAL CORONARY ATHERECTOMY, WITH INTRACORONARY STENT, WITH CORONARY ANGIOPLASTY WHEN | |
| History of surgical or PERFORMED; EACH ADDITIONAL BRANCH OF A MAJOR CORONARY | |
| percutaneous coronary ARTERY (LIST SEPARATELY IN ADDITION TO CODE FOR PRIMARY | |
| <b>4.1.4</b> revascularization procedure 92934 PX PROCEDURE) ICD-1 | 0-PCS |


PERCUTANEOUS TRANSLUMINAL REVASCULARIZATION OF OR


TRANSCATHETER PLACEMENT OF AN INTRAVASCULAR STENT(S)


Component 1 overlap with component 2 OR component 3


TRANSCATHETER AORTIC VALVE REPLACEMENT (TAVR/TAVI) WITH


| Bariatric surgery within 13 the past 12 months | 43846 PX | GASTRIC RESTRICTIVE PROCEDURE, WITH GASTRIC BYPASS, FOR MORBID OBESITY; WITH SHORT LIMB (LESS THAN 100 CM) ROUX-EN-Y GASTROENTEROSTOMY | CPT/HCPCS |
|---|---|---|---|
| Bariatric surgery within | | GASTRIC RESTRICTIVE PROCEDURE, WITH SMALL INTESTINE RECONSTRUCTION | I |
| 13 the past 12 months Bariatric surgery within | 43847 PX | TO LIMIT ABSORPTION; WITH LONG LIMB (>150 CM) ROUX-EN-Y GASTRECTOMY, TOTAL; WITH ROUX-EN-Y RECONSTRUCTION; MINI-GASTRIC | CPT/HCPCS |
| 13 the past 12 months Bariatric surgery within | 43659 PX | BYPASS<br>LAPAROSCOPY, SURGICAL; GASTRIC RESTRICTIVE PROCEDURE, ADJUSTABLE | CPT/HCPCS |
| 13 the past 12 months Bariatric surgery within | S2082 PX | GASTRIC BAND INCLUDES PLACEMENT OF SUBCUTANEOUS PORT | CPT/HCPCS |
| 13 the past 12 months Bariatric surgery within | S2085 PX | LAPAROSCOPIC GASTRIC BYPASS LAPAROSCOPY, SURGICAL, GASTRIC RESTRICTIVE PROCEDURE: LONGITUDINAL | CPT/HCPCS |
| 13 the past 12 months Bariatric surgery within | 43775 PX | GASTRECTOMY (E.G., SLEEVE GASTRECTOMY) | CPT/HCPCS |
| 13 the past 12 months | 43848 PX | REVISION RYGB | CPT/HCPCS |


CEREBRAL INFARCTION DUE TO THROMBOSIS


CEREBRAL INFARCTION DUE TO EMBOLISM OF


OCCLUSION AND STENOSIS OF UNSPECIFIED


In combination with intravenous administration In combination with intravenous administration In combination with intravenous administration

In combination with intravenous administration

In combination with intravenous administration In combination with generic drug name codes for furosemide, torsemide, bumetanide


N/A

N/A N/A N/A

Codes indicate stage V or endstage renal disease (ESRD)

#### Appendix 3. Flowchart for cohort assembly

| OPTUM (May 13, 2022 to Feb 28, 2025) | | |
|---|---|---|
| | Excluded Patients | Remaining Patients |
| Patients in dataset | | 95,349,41 |
| Patients meeting cohort entry criteria | | 916,84 |
| Excluded due to insufficient enrollment | -321,216 (35%) | 595,63 |
| Excluded due to prior use of referent | -240,911 (40%) | 354,72 |
| Excluded due to prior use of exposure | -117,929 (33%) | 236,79 |
| Excluded because patient qualified in >1 exposure category | -7 (<1%) | 236,784 |
| Excluded based on 1 - Age | -78 (<1%) | 236,706 |
| Excluded based on 1 - Gender | -18 (<1%) | 236,688 |
| Excluded based on 2 - Type 2 diabetes mellitus | -16,091 (7%) | 220,59 |
| Excluded based on 3 - BMI ≥ 25kg/m2 (ICD-10) | -17,972 (8%) | 202,625 |
| Excluded based on 3 - BMI ≥ 25kg/m2 (Truncated) | -485 (<1%) | 202,140 |
| Excluded based on 4 - Increased cardiovascular risk | -2,482 (1%) | 199,658 |
| Excluded based on 5 - History of T1DM or secondary diabetes | -1,800 (<1%) | 197,858 |
| Excluded based on 6 - Family or personal history of multiple endocrine neoplasia or medullary thyroid carcinoma | -258 (<1%) | 197,60 |
| Excluded based on 7 - End-stage renal disease or dialysis | -885 (<1%) | 196,71 |
| Excluded based on 8 - History of treatment for diabetic retinopathy and/or macular edema | -1,263 (<1%) | 195,45 |
| Excluded based on 9 - History of any malignancy | -5,377 (3%) | 190,07 |
| Excluded based on 10 - Cardiovascular event or intervention in the past 7 days | -69 (<1%) | 190,000 |
| Excluded based on 11 - Women who are pregnant or breastfeeding | -67 (<1%) | 189,93 |
| Excluded based on 12 - GLP-1-RA treatment within past 6 months | -3,554 (2%) | 186,38 |
| Excluded based on 13 - Bariatric surgery within the past 12 months | -524 (<1%) | 185,86 |
| Patients in Exposure Group | | 61,22 |
| Patients in Referent Group | | 124,63 |
| Total Patients | | 185.86 |

| | Excluded Patients | Remaining Patients |
|---|---|---|
| Patients in dataset | | 126,118,01 |
| Patients meeting cohort entry criteria | | 658,159 |
| Excluded due to insufficient enrollment | -125,338 (19%) | 532,82 |
| Excluded due to prior use of referent | -293,040 (55%) | 239,78 |
| Excluded due to prior use of exposure | -85,822 (36%) | 153,959 |
| Excluded because patient qualified in >1 exposure category | -9 (<1%) | 153,950 |
| Excluded based on 1 - Age | -231 (<1%) | 153,719 |
| Excluded based on 1 - Gender | -0 (<1%) | 153,719 |
| Excluded based on 2 - Type 2 diabetes mellitus | -37,200 (24%) | 116,519 |
| Excluded based on 3 - BMI ≥ 25kg/m2 (ICD-10) | -11,742 (10%) | 104,77 |
| Excluded based on 4 - Increased cardiovascular risk | -2,907 (3%) | 101,870 |
| Excluded based on 5 - History of T1DM or secondary diabetes | -964 (<1%) | 100,906 |
| Excluded based on 6 - Family or personal history of multiple endocrine neoplasia or medullary thyroid carcinoma | -167 (<1%) | 100,73 |
| Excluded based on 7 - End-stage renal disease or dialysis | -257 (<1%) | 100,48 |
| Excluded based on 8 - History of treatment for diabetic retinopathy and/or macular edema | -457 (<1%) | 100,029 |
| Excluded based on 9 - History of any malignancy | -2,167 (2%) | 97,858 |
| Excluded based on 10 - Cardiovascular event or intervention in the past 7 days | -39 (<1%) | 97,819 |
| Excluded based on 11 - Women who are pregnant or breastfeeding | -131 (<1%) | 97,688 |
| Excluded based on 12 - GLP-1-RA treatment within past 6 months | -3,036 (3%) | 94,65 |
| Excluded based on 13 - Bariatric surgery within the past 12 months | -291 (<1%) | 94,36 |
| Patients in Exposure Group | | 25,384 |
| Patients in Referent Group | | 68,97 |
| Total Patients | | 94.36 |

#### Appendix 4.1st Feasibility Assessment

#### Table of Contents

- A. Patient characteristics by treatment group
- B. Summary Parameters of Study Population
- C. Median Follow up Time in Overall Study Population
- D. Reasons for Censoring in Overall Study Population
- E. Initial Power Assessment
- F. Aetion report link
- G. Review by Principal Investigator

In order to complete the initial power analysis, a dummy outcome of a 90-day gap in database enrollment was used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. We completed a PS overlap weighted comparative analysis using this outcome. The PS included only 3 covariates: age, sex, and combined comorbidity index. Power calculations are based on the formulas from Chow et al. (2008).

OPTUM: Study period from May 13, 2022 to Feb 28, 2025 MARKETSCAN: Study period from May 13, 2022 to Dec 31, 2023

### A. Patient characteristics by treatment group (follow-up start is 1 days after CED, so few patients and dropped, hence table 1 could include sightly fewer patients than the attrition table)

| Before matching | | Optum | | Marketscan | | |
|---|---|---|---|---|---|---|
| Variable | Exposure: Semaglutide injection | Exposure: Tirzepatide | Difference | Exposure: Semaglutide injection | Exposure: Tirzepatide | Difference |
| Number of patients | 124,634 | 61,227 | - (-, -) | 68,977 | 25,384 | - (-, -) |
| Age | | | | | | |
| mean (sd) | 63.53 (11.03) | 61.45 (11.51) | 2.08 (1.97, 2.19) | 54.47 (10.20) | 53.78 (9.96) | 0.68 (0.54, 0.83) |
| median [IQR] | 66.00 [56.00, 71.00] | 63.00 [54.00, 70.00] | - (-, -) | 55.00 [48.00, 61.00] | 54.00 [48.00, 60.00] | - (-, -) |
| Gender | | | | | | |
| Male; n (%) | 54,169 (43.5%) | 27,096 (44.3%) | -0.8% (-1.3%, -0.3%) | 30,813 (44.7%) | 11,256 (44.3%) | 0.3% (-0.4%, 1.0%) |
| CCI (365 days) | | | | | | |
| mean (sd) | 2.00 (2.40) | 1.79 (2.27) | 0.21 (0.19, 0.24) | 0.98 (1.67) | 0.92 (1.57) | 0.06 (0.04, 0.08) |
| median [IQR] | 1.00 [0.00, 3.00] | 1.00 [0.00, 3.00] | - (-, -) | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | - (-, -) |

#### B. Summary Parameters of Overall Study Population (Step 1)

| | Optum | Marketscan |
|-----------------------------------------------------|-----------|------------|
| Variable | Value | Value |
| Number of patients in full cohort | 185,861 | 94,361 |
| Number of patients dropped as incomplete cases | 0 | 0 |
| Number of patients that did not begin follow-up | 299 | 72 |
| Number of patients in analytic cohort | 185,562 | 94,289 |
| Number of events | 1,699 | 347 |
| Number of person-years | 93,424.06 | 42,930.20 |
| Number of patients in group: Reference-Sitagliptin | 124,470 | 68,932 |
| Number of patients in group: Exposure - Tirzepatide | 61,092 | 25,357 |
| Risk per 1,000 patients | 9.16 | 3.68 |
| Rate per 1,000 person-years | 18.19 | 8.08 |

### C. Median Follow up Time in Overall Study Population (Step 1)

| | Optum | Marketscan |
|----------------------------|------------------------------|------------------|
| Patient Group | Median Follow-Up Time (Days) | Median Follow-Up |
| Overall Patient Population | 154 [85, 286] | 143 [73, 243] |

## D. Reasons for Censoring in Overall Study Population (Step 1)

| | Optum | Marketscan |
|---|---|---|
| Overall | Value | Value |
| Outcome | 1,699 (0.9%) | 347 (0.4%) |
| Start of an additional exposure | 7,362 (4.0%) | 3,572 (3.8%) |
| End of index exposure | 74,779 (40.3%) | 27,446 (29.1%) |
| Maximum follow-up time | 31,515 (17.0%) | 8,157 (8.7%) |
| Specified date reached | 14,608 (7.9%) | 46,266 (49.1%) |
| End of patient data | 0 (0.0%) | 0 (0.0%) |
| End of patient enrollment | 50,722 (27.3%) | 6,186 (6.6%) |
| Switch to other GLP-1-RA (for censoring) / Nursing home admission | 4,877 (2.6%) | 2,315 (2.5%) |

### E. Power Assessment

| Noninferiority Analysis | Optum | Marketscan |
|----------------------------|---------|------------|
| Number of patients matched | | |
| Reference | 124,634 | 68,977 |
| Exposed | 61,227 | 25,384 |
| Risk per 1,000 patients | 9.16 | 3.68 |
| Assumed HR from RCT | 0.9 | 0.9 |
| Alpha (2-sided) | 0.05 | 0.05 |
| Non-inferiority margin | 1.05 | 1.05 |
| Number of events expected | 1702 | 347 |
| Power | 0.89 | 0.30 |

### F. Aetion report link

Optum Step 1: https://bwh-dopeaetion.com/project/2916/rwrs/139403 Marketscan Step 1: https://bwh-dopeaetion.com/project/2915/rwrs/139405

## F. Review by principal investigator

Stop analyses until feasibility and power are reviewed by primary investigators.

| Reviewed by PI: | Nils Krüger | Date reviewed: | July 30, 2025 |
|-----------------|-------------|----------------|---------------|

# Appendix 5. 2nd Feasibility Assessment

### **Table of Contents**

A. Median Follow up Time by Treatment Group

B. Reasons for Censoring by Treatment Group

C. Final Power Assessment

D. Aetion report link

E. Review by Principal Investigator

In order to complete the feasibility analysis, a dummy outcome of a 90-day gap in database enrollment was used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. We completed a PS overlap weighted comparative analysis using this outcome. The PS included all prespecified covariates listed in the protocol. Power calculations are based on the

# A. Median Follow Up Time by Treatment Group

| Patient Group | • | Median Follow-Up<br>Time (Days) [IQR] |
|---|---|---|
| Overall Patient Population | 154 [85, 286] | 143 [73, 243] |

# B. Reasons for Censoring in Overall Study Population

| | Optum | Marketscan |
|---|---|---|
| Overall | Value | Value |
| Outcome | 1,699 (0.9%) | 347 (0.4%) |
| Start of an additional exposure | 7,362 (4.0%) | 3,572 (3.8%) |
| End of index exposure | 74,779 (40.3%) | 27,446 (29.1%) |
| Maximum follow-up time | 31,515 (17.0%) | 8,157 (8.7%) |
| Specified date reached | 14,608 (7.9%) | 46,266 (49.1%) |
| End of patient data | 0 (0.0%) | 0 (0.0%) |
| End of patient enrollment | 50,722 (27.3%) | 6,186 (6.6%) |
| Switch to other GLP-1-RA (for censoring) / Nursing home admission | 4,877 (2.6%) | 2,315 (2.5%) |

## **C. Power Assessment**

| Noninferiority Analysis | Optum | Marketscan |
|----------------------------|---------|------------|
| Number of patients matched | | |
| Reference | 124,634 | 68,977 |
| Exposed | 61,227 | 25,384 |
| Risk per 1,000 patients | 9.16 | 3.68 |
| Assumed HR from RCT | 0.9 | 0.9 |
| Alpha (2-sided) | 0.05 | 0.05 |

| Non-inferiority margin | 1.05 | 1.05 |
|---------------------------|------|------|
| Number of events expected | 1702 | 347 |
| Power | 0.89 | 0.30 |

# D. Aetion report link

Optum Step 1: https://bwh-dope.aetion.com/project/2916/rwrs/139403 Marketscan Step 1: https://bwh-dope.aetion.com/project/2915/rwrs/139405

# E. Review by principal investigator

Stop analyses until feasibility and power are reviewed by primary investigators.

| Reviewed by PI: | Nils Krüger | Date reviewed: | July 30, 2025 |
|-----------------|-------------|----------------|---------------|

### Appendix 6. Balance Assessment - PS Distribution and C-Statistic





### C-statistics adjusted after overlap weighing on the PS, OPTUM: 0.511



### C-statistics unadjusted, MARKETSCAN: 0.603



### C-statistics adjusted after overlap weighing on the PS, MARKETSCAN: 0.518



Appendix 7. Balance Assessment - Table 1

| ОРТИМ | T T | | | 1 | | |
|---|---|---|---|---|---|---|
| Variable | Exposure: Semaglutide injection | Exposure: Tirzepatide | Difference | Exposure: Semaglutide injection | Exposure: Tirzepatide | Difference |
| Number of patients | 124,470 | 61,092 | - (-, -) | 60,848 | 60,848 | - (-, -) |
| Year of Cohort Entry Date | 124,470 | 61,032 | - (-, -) | 60,848 | 60,046 | - (-, -) |
| 2022: n (%) | 19.394 (15.6%) | 5.376 (8.8%) | 6.8% (6.5%, 7.1%) | 5.211 (8.6%) | 5.376 (8.8%) | -0.3% (-0.6%, 0.0%) |
| 2023; n (%) | 51,514 (41.4%) | 24,848 (40.7%) | 0.7% (0.2%, 1.2%) | 25,051 (41.2%) | 24,830 (40.8%) | 0.4% (-0.2%, 0.9%) |
| 2024; n (%) | 52.184 (41.9%) | 29,476 (48.2%) | -6.3% (-6.8%, -5.8%) | 29,373 (48.3%) | 29,379 (48.3%) | -0.0% (-0.6%, 0.6%) |
| 2025; n (%) | 1,378 (1.1%) | 1,392 (2.3%) | -1.2% (-1.3%, -1.0%) | 1,213 (2.0%) | 1,263 (2.1%) | -0.1% (-0.2%, 0.1%) |
| Age | 1,070 (1170) | 1,002 (L.O70) | 11270 ( 11070, 11070) | 1,210 (2.070) | 1,200 (2,170) | 0.270 ( 0.270, 0.270) |
| mean (sd) | 63.53 (11.03) | 61.44 (11.51) | 2.09 (1.98, 2.20) | 61.51 (11.60) | 61.51 (11.46) | -0.01 (-0.14, 0.12) |
| median [IQR] | 66.00 [56.00, 71.00] | 63.00 [54.00, 70.00] | - (-, -) | 64.00 [54.00, 70.00] | 64.00 [54.00, 70.00] | - (-, -) |
| min, max | 18.00, 88.00 | 18.00, 88.00 | - (-, -) | 18.00, 88.00 | 18.00, 88.00 | - (-, -) |
| Gender (male); n (%) | 54,100 (43.5%) | 27,036 (44.3%) | -0.8% (-1.3%, -0.3%) | 27,058 (44.5%) | 26,924 (44.2%) | 0.2% (-0.3%, 0.8%) |
| Race (Recategorized) | | , | | | | |
| White; n (%) | 56,020 (45.0%) | 27,751 (45.4%) | -0.4% (-0.9%, 0.1%) | 27,719 (45.6%) | 27,636 (45.4%) | 0.1% (-0.4%, 0.7%) |
| Black; n (%) | 17,194 (13.8%) | 7,565 (12.4%) | 1.4% (1.1%, 1.8%) | 7,544 (12.4%) | 7,550 (12.4%) | -0.0% (-0.4%, 0.4%) |
| Unknown / Missing; n (%) | 49,204 (39.5%) | 24,906 (40.8%) | -1.2% (-1.7%, -0.8%) | 24,731 (40.6%) | 24,793 (40.7%) | -0.1% (-0.7%, 0.5%) |
| Others; n (%) | 2,052 (1.6%) | 870 (1.4%) | 0.2% (0.1%, 0.3%) | 854 (1.4%) | 869 (1.4%) | -0.0% (-0.2%, 0.1%) |
| Region / State | | | | | | |
| Northest; n (%) | 11,459 (9.2%) | 4,598 (7.5%) | 1.7% (1.4%, 1.9%) | 4,586 (7.5%) | 4,597 (7.6%) | -0.0% (-0.3%, 0.3%) |
| Midwest / North central; n (%) | 25,578 (20.5%) | 13,148 (21.5%) | -1.0% (-1.4%, -0.6%) | 13,149 (21.6%) | 13,108 (21.5%) | 0.1% (-0.4%, 0.5%) |
| South; n (%) | 66,847 (53.7%) | 35,371 (57.9%) | -4.2% (-4.7%, -3.7%) | 35,105 (57.7%) | 35,174 (57.8%) | -0.1% (-0.7%, 0.4%) |
| West; n (%) | 20,534 (16.5%) | 7,938 (13.0%) | 3.5% (3.2%, 3.8%) | 7,973 (13.1%) | 7,933 (13.0%) | 0.1% (-0.3%, 0.4%) |
| Missing; n (%) | 52 (0.0%) | 37 (0.1%) | -0.0% (-0.0%, 0.0%) | 35 (0.1%) | 36 (0.1%) | -0.0% (-0.0%, 0.0%) |
| Smoking/Tobacco use; n (%) | 30,627 (24.6%) | 13,928 (22.8%) | 1.8% (1.4%, 2.2%) | 13,880 (22.8%) | 13,887 (22.8%) | -0.0% (-0.5%, 0.5%) |
| Weight | | | | | | |
| Overweight; n (%) | 9,152 (7.4%) | 3,744 (6.1%) | 1.2% (1.0%, 1.5%) | 3,694 (6.1%) | 3,743 (6.2%) | -0.1% (-0.4%, 0.2%) |
| Class 1 Obesity; n (%) | 24,459 (19.7%) | 10,774 (17.6%) | 2.0% (1.6%, 2.4%) | 10,770 (17.7%) | 10,753 (17.7%) | 0.0% (-0.4%, 0.5%) |
| Class 2 Obesity; n (%) | 38,113 (30.6%) | 18,929 (31.0%) | -0.4% (-0.8%, 0.1%) | 18,980 (31.2%) | 18,869 (31.0%) | 0.2% (-0.3%, 0.7%) |
| Class 3 Obesity; n (%) | 34,833 (28.0%) | 18,995 (31.1%) | -3.1% (-3.6%, -2.7%) | 18,783 (30.9%) | 18,854 (31.0%) | -0.1% (-0.6%, 0.4%) |
| Unspecified Obesity; n (%) | 17,913 (14.4%) | 8,650 (14.2%) | 0.2% (-0.1%, 0.6%) | 8,621 (14.2%) | 8,629 (14.2%) | -0.0% (-0.4%, 0.4%) |
| Diabetic retinopathy; n (%) | 10,581 (8.5%) | 4,649 (7.6%) | 0.9% (0.6%, 1.2%) | 4,648 (7.6%) | 4,648 (7.6%) | 0.0% (-0.3%, 0.3%) |
| Diabetic neuropathy; n (%) | 32,680 (26.3%) | 14,434 (23.6%) | 2.6% (2.2%, 3.0%) | 14,224 (23.4%) | 14,413 (23.7%) | -0.3% (-0.8%, 0.2%) |
| Diabetic nephropathy; n (%) | 27,397 (22.0%) | 11,637 (19.0%) | 3.0% (2.6%, 3.4%) | 11,587 (19.0%) | 11,622 (19.1%) | -0.1% (-0.5%, 0.4%) |
| Diabetes with other ophthalmic complications; n (%) | 5,448 (4.4%) | 2,138 (3.5%) | 0.9% (0.7%, 1.1%) | 2,082 (3.4%) | 2,135 (3.5%) | -0.1% (-0.3%, 0.1%) |
| Diabetes with peripheral circulatory disorders; n (%) | 18,230 (14.6%) | 7,894 (12.9%) | 1.7% (1.4%, 2.1%) | 7,929 (13.0%) | 7,883 (13.0%) | 0.1% (-0.3%, 0.5%) |
| Diabetic foot; n (%) | 3,638 (2.9%) | 1,652 (2.7%) | 0.2% (0.1%, 0.4%) | 1,609 (2.6%) | 1,650 (2.7%) | -0.1% (-0.3%, 0.1%) |
| Erectile dysfunction; n (%) | 6,091 (4.9%) | 3,050 (5.0%) | -0.1% (-0.3%, 0.1%) | 3,073 (5.1%) | 3,038 (5.0%) | 0.1% (-0.2%, 0.3%) |
| Hypoglycemia; n (%) | 31,299 (25.1%) | 14,971 (24.5%) | 0.6% (0.2%, 1.1%) | 14,869 (24.4%) | 14,920 (24.5%) | -0.1% (-0.6%, 0.4%) |
| Hyperglycemia/DKA/HONK; n (%) | 61,623 (49.5%) | 30,454 (49.8%) | -0.3% (-0.8%, 0.1%) | 30,179 (49.6%) | 30,310 (49.8%) | -0.2% (-0.8%, 0.3%) |
| Skin infections; n (%) | 12,767 (10.3%) | 6,441 (10.5%) | -0.3% (-0.6%, 0.0%) | 6,325 (10.4%) | 6,397 (10.5%) | -0.1% (-0.5%, 0.2%) |
| Stable angina; n (%) | 6,228 (5.0%) | 2,606 (4.3%) | 0.7% (0.5%, 0.9%) | 2,619 (4.3%) | 2,604 (4.3%) | 0.0% (-0.2%, 0.3%) |
| Unstable angina; n (%) | 3,044 (2.4%) | 1,325 (2.2%) | 0.3% (0.1%, 0.4%) | 1,328 (2.2%) | 1,323 (2.2%) | 0.0% (-0.2%, 0.2%) |
| Hypertension; n (%) | 110,340 (88.6%) | 53,374 (87.4%) | 1.3% (1.0%, 1.6%) | 53,205 (87.4%) | 53,180 (87.4%) | 0.0% (-0.3%, 0.4%) |
| Hypotension; n (%) | 3,805 (3.1%) | 1,648 (2.7%) | 0.4% (0.2%, 0.5%) | 1,586 (2.6%) | 1,646 (2.7%) | -0.1% (-0.3%, 0.1%) |
| Hyperlipidemia; n (%) | 106,301 (85.4%) | 51,835 (84.8%) | 0.6% (0.2%, 0.9%) | 51,546 (84.7%) | 51,642 (84.9%) | -0.2% (-0.6%, 0.2%) |
| Atrial fibrillation; n (%) | 12,842 (10.3%) | 5,568 (9.1%) | 1.2% (0.9%, 1.5%) | 5,545 (9.1%) | 5,557 (9.1%) | -0.0% (-0.3%, 0.3%) |
| Cardiac conduction disorder; n (%) | 7,504 (6.0%) | 3,180 (5.2%) | 0.8% (0.6%, 1.0%) | 3,216 (5.3%) | 3,175 (5.2%) | 0.1% (-0.2%, 0.3%) |
| Previous cardiac procedure (CABG, PTCA, Stent); n (%) | 2,068 (1.7%) | 800 (1.3%) | 0.4% (0.2%, 0.5%) | 813 (1.3%) | 800 (1.3%) | 0.0% (-0.1%, 0.2%) |
| Ischemic stroke; n (%) | 835 (0.7%) | 285 (0.5%) | 0.2% (0.1%, 0.3%) | 274 (0.5%) | 285 (0.5%) | -0.0% (-0.1%, 0.1%) |
| PVD diagnosis or surgery; n (%) | 12,113 (9.7%) | 5,100 (8.3%) | 1.4% (1.1%, 1.7%) | 5,027 (8.3%) | 5,096 (8.4%) | -0.1% (-0.4%, 0.2%) |
| Other cardiac dysrhythmia; n (%) | 25,863 (20.8%) | 11,891 (19.5%) | 1.3% (0.9%, 1.7%)<br>0.9% (0.6%, 1.1%) | 11,830 (19.4%) | 11,846 (19.5%) | -0.0% (-0.5%, 0.4%) |
| Cardiomyopathy; n (%) | 6,554 (5.3%) | 2,695 (4.4%) | | 2,730 (4.5%) | 2,694 (4.4%) | 0.1% (-0.2%, 0.3%) |
| Valve disorders; n (%) | 13,800 (11.1%)<br>1,510 (1.2%) | 6,049 (9.9%)<br>605 (1.0%) | 1.2% (0.9%, 1.5%)<br>0.2% (0.1%, 0.3%) | 6,035 (9.9%)<br>621 (1.0%) | 6,044 (9.9%)<br>605 (1.0%) | -0.0% (-0.4%, 0.3%)<br>0.0% (-0.1%, 0.1%) |
| Valve replacement; n (%) TIA; n (%) | 2,172 (1.7%) | 887 (1.5%) | 0.2% (0.1%, 0.3%) | 905 (1.5%) | 885 (1.5%) | 0.0% (-0.1%, 0.1%) |
| | 2,172 (1.7%)<br>17,517 (14.1%) | 8,277 (13.5%) | 0.5% (0.2%, 0.4%) | 8,154 (13.4%) | 8,249 (13.6%) | -0.2% (-0.5%, 0.2%) |
| Edema; n (%) Venous thromboembolism / Pulmonary embolism; n (%) | 4,042 (3.2%) | 8,277 (13.5%)<br>1.917 (3.1%) | 0.5% (0.2%, 0.9%) | 1.882 (3.1%) | 1.907 (3.1%) | -0.2% (-0.5%, 0.2%) |
| Venous thromboembolism / Pulmonary embolism; n (%) Pulmonary hypertension; n (%) | 4,042 (3.2%) 4,009 (3.2%) | 1,917 (3.1%) 1,736 (2.8%) | 0.1% (-0.1%, 0.3%) | 1,769 (2.9%) | 1,907 (3.1%)<br>1,734 (2.8%) | -0.0% (-0.2%, 0.2%)<br>0.1% (-0.1%, 0.2%) |
| Pulmonary nypertension; n (%) Implantable cardioverter defibrillator; n (%) | 4,009 (3.2%)<br>299 (0.2%) | 1,736 (2.8%) | -0.0% (-0.1%, 0.0%) | 1,769 (2.9%) 158 (0.3%) | 1,734 (2.8%) | 0.1% (-0.1%, 0.2%) |
| Implantable cardioverter defibrillator; n (%) Hyperkalemia; n (%) | 3,888 (3.1%) | 1,527 (2.5%) | -0.0% (-0.1%, 0.0%)<br>0.6% (0.5%, 0.8%) | 1,493 (2.5%) | 151 (0.2%)<br>1,525 (2.5%) | -0.1% (-0.2%, 0.1%) |
| нурегканетна; n (%) Coronary atherosclerosis; n (%) | 27,304 (21.9%) | 1,527 (2.5%) | 2.3% (1.9%, 2.7%) | 1,493 (2.5%) 12,009 (19.7%) | 1,525 (2.5%) 11,965 (19.7%) | 0.1% (-0.2%, 0.1%) |
| Coronary atheroscierosis; n (%) Cerebrovascular procedure: n (%) | 27,304 (21.9%)<br>172 (0.1%) | 11,979 (19.6%)<br>55 (0.1%) | 0.0% (0.0%, 0.1%) | 12,009 (19.7%)<br>56 (0.1%) | 11,965 (19.7%)<br>55 (0.1%) | 0.1% (-0.4%, 0.5%) |
| | 220 (0.2%) | 89 (0.1%) | 0.0% (0.0%, 0.1%) | 92 (0.2%) | 89 (0.1%) | 0.0% (-0.0%, 0.0%) |
| Insertion of pacemakers / removal of cardiac lead; n (%) | ZZU (U.Z70) | 03 (0.1%) | U.U70 (-U.U%, U.1%) | JZ (U.Z70) | OJ (U.1%) | U.U70 (-U.U70, U.U70) |

| CKD Stage 1-2; n (%) | 6,855 (5.5%) | 3,008 (4.9%) | 0.6% (0.4%, 0.8%) | 2,986 (4.9%) | 3,003 (4.9%) | -0.0% (-0.3%, 0.2%) |
|---|---|---|---|---|---|---|
| CKD Stage 3-4; n (%) | 20,201 (16.2%) | 8,251 (13.5%) | 2.7% (2.4%, 3.1%) | 8,173 (13.4%) | 8,247 (13.6%) | -0.1% (-0.5%, 0.3%) |
| Unspecified CKD; n (%) | 7,809 (6.3%) | 3,127 (5.1%) | 1.2% (0.9%, 1.4%) | 3,059 (5.0%) | 3,125 (5.1%) | -0.1% (-0.4%, 0.1%) |
| Acute kidney injury; n (%) | 7,820 (6.3%) | 3,127 (5.1%) | 1.2% (0.9%, 1.4%) | 3,107 (5.1%) | 3,125 (5.1%) | -0.0% (-0.3%, 0.2%) |
| Hypertensive nephropathy; n (%) | 16,767 (13.5%) | 6,778 (11.1%) | 2.4% (2.1%, 2.7%) | 6,719 (11.0%) | 6,775 (11.1%) | -0.1% (-0.4%, 0.3%) |
| Urinary tract infections; n (%) | 16,712 (13.4%) | 7,787 (12.7%) | 0.7% (0.4%, 1.0%) | 7,633 (12.5%) | 7,766 (12.8%) | -0.2% (-0.6%, 0.2%) |
| Genital infections; n (%) | 3,779 (3.0%) | 1,724 (2.8%) | 0.2% (0.1%, 0.4%) | 1,708 (2.8%) | 1,715 (2.8%) | -0.0% (-0.2%, 0.2%) |
| Urolithiasis (Kidney and urinary stone); n (%) | 5,842 (4.7%) | 2,818 (4.6%) | 0.1% (-0.1%, 0.3%) | 2,818 (4.6%) | 2,807 (4.6%) | 0.0% (-0.2%, 0.3%) |
| COPD; n (%) | 16,510 (13.3%) | 6,932 (11.3%) | 1.9% (1.6%, 2.2%) | 6,952 (11.4%) | 6,932 (11.4%) | 0.0% (-0.3%, 0.4%) |
| Asthma; n (%) | 16,060 (12.9%) | 7,806 (12.8%) | 0.1% (-0.2%, 0.5%) | 7,774 (12.8%) | 7,779 (12.8%) | -0.0% (-0.4%, 0.4%) |
| Obstructive sleep apnea; n (%) | 40,962 (32.9%) | 20,912 (34.2%) | -1.3% (-1.8%, -0.9%) | 20,789 (34.2%) | 20,821 (34.2%) | -0.1% (-0.6%, 0.5%) |
| Serious bacterial infections; n (%) | 3,364 (2.7%) | 1,464 (2.4%) | 0.3% (0.2%, 0.5%) | 1,398 (2.3%) | 1,462 (2.4%) | -0.1% (-0.3%, 0.1%) |
| Pneumonia: n (%) | 5.894 (4.7%) | 2.495 (4.1%) | 0.7% (0.5%, 0.8%) | 2.535 (4.2%) | 2,491 (4.1%) | 0.1% (-0.2%, 0.3%) |
| Liver disease; n (%) | 22,532 (18.1%) | 11,110 (18.2%) | -0.1% (-0.5%, 0.3%) | 11,028 (18.1%) | 11,042 (18.1%) | -0.0% (-0.5%, 0.4%) |
| MASH/MASLD; n (%) | 12,872 (10.3%) | 6,897 (11.3%) | -0.9% (-1.3%, -0.6%) | 6,853 (11.3%) | 6,838 (11.2%) | 0.0% (-0.3%, 0.4%) |
| Fractures / Falls; n (%) | 7,543 (6.1%) | 3,367 (5.5%) | 0.5% (0.3%, 0.8%) | 3,339 (5.5%) | 3,358 (5.5%) | -0.0% (-0.3%, 0.2%) |
| Osteoporosis; n (%) | 5,807 (4.7%) | 2,412 (3.9%) | 0.7% (0.5%, 0.9%) | 2,363 (3.9%) | 2,412 (4.0%) | -0.1% (-0.3%, 0.1%) |
| Osteoarthritis; n (%) | 39,976 (32.1%) | 18,495 (30.3%) | 1.8% (1.4%, 2.3%) | 18,480 (30.4%) | 18,468 (30.4%) | 0.0% (-0.5%, 0.5%) |
| | 27,794 (22.3%) | 13,102 (21.4%) | 0.9% (0.5%, 1.3%) | 13,073 (21.5%) | 13,048 (21.4%) | 0.0% (-0.4%, 0.5%) |
| Depression; n (%) | | | | | | |
| Dementia; n (%) | 4,092 (3.3%) | 1,508 (2.5%) | 0.8% (0.7%, 1.0%) | 1,416 (2.3%) | 1,507 (2.5%) | -0.1% (-0.3%, 0.0%) |
| Delirium or psychosis; n (%) | 2,150 (1.7%) | 789 (1.3%) | 0.4% (0.3%, 0.6%) | 776 (1.3%) | 788 (1.3%) | -0.0% (-0.1%, 0.1%) |
| Anxiety; n (%) | 29,246 (23.5%) | 14,681 (24.0%) | -0.5% (-0.9%, -0.1%) | 14,618 (24.0%) | 14,607 (24.0%) | 0.0% (-0.5%, 0.5%) |
| Sleep disorders; n (%) | 44,883 (36.1%) | 21,940 (35.9%) | 0.1% (-0.3%, 0.6%) | 21,784 (35.8%) | 21,852 (35.9%) | -0.1% (-0.7%, 0.4%) |
| Anemia; n (%) | 23,303 (18.7%) | 10,777 (17.6%) | 1.1% (0.7%, 1.5%) | 10,700 (17.6%) | 10,738 (17.6%) | -0.1% (-0.5%, 0.4%) |
| Influenza; n (%) | 2,349 (1.9%) | 1,327 (2.2%) | -0.3% (-0.4%, -0.1%) | 1,270 (2.1%) | 1,317 (2.2%) | -0.1% (-0.2%, 0.1%) |
| COVID; n (%) | 13,619 (10.9%) | 6,549 (10.7%) | 0.2% (-0.1%, 0.5%) | 6,414 (10.5%) | 6,528 (10.7%) | -0.2% (-0.5%, 0.2%) |
| Hyperthyroidism and other thyroid gland disorders; n (%) | 32,597 (26.2%) | 16,115 (26.4%) | -0.2% (-0.6%, 0.2%) | 15,985 (26.3%) | 16,048 (26.4%) | -0.1% (-0.6%, 0.4%) |
| Hypothyroidism; n (%) | 26,425 (21.2%) | 13,037 (21.3%) | -0.1% (-0.5%, 0.3%) | 12,936 (21.3%) | 12,988 (21.3%) | -0.1% (-0.5%, 0.4%) |
| Nephrotic syndrome; n (%) | 107 (0.1%) | 49 (0.1%) | 0.0% (-0.0%, 0.0%) | 46 (0.1%) | 48 (0.1%) | -0.0% (-0.0%, 0.0%) |
| Urinary incontinence; n (%) | 7,488 (6.0%) | 3,265 (5.3%) | 0.7% (0.4%, 0.9%) | 3,201 (5.3%) | 3,259 (5.4%) | -0.1% (-0.3%, 0.2%) |
| Biliary disease; n (%) | 161 (0.1%) | 71 (0.1%) | 0.0% (-0.0%, 0.0%) | 67 (0.1%) | 71 (0.1%) | -0.0% (-0.0%, 0.0%) |
| Pancreatitis; n (%) | 125 (0.1%) | 57 (0.1%) | 0.0% (-0.0%, 0.0%) | 70 (0.1%) | 57 (0.1%) | 0.0% (-0.0%, 0.1%) |
| Bowel obstruction; n (%) | 132 (0.1%) | 77 (0.1%) | -0.0% (-0.1%, 0.0%) | 75 (0.1%) | 76 (0.1%) | -0.0% (-0.0%, 0.0%) |
| Gastroparesis: n (%) | 989 (0.8%) | 573 (0.9%) | -0.1% (-0.2%, -0.1%) | 548 (0.9%) | 562 (0.9%) | -0.0% (-0.1%, 0.1%) |
| Gastroparesis; n (%) Number of antidiabetic drugs on CED | 989 (0.8%) | 573 (0.9%) | -0.1% (-0.2%, -0.1%) | 548 (0.9%) | 562 (0.9%) | -0.0% (-0.1%, 0.1%) |
| Number of antidiabetic drugs on CED | · | | | | | |
| Number of antidiabetic drugs on CEDmean (sd) | 2.12 (0.96) | 2.08 (0.96) | 0.04 (0.03, 0.05) | 2.08 (0.95) | 2.08 (0.96) | -0.00 (-0.01, 0.01) |
| Number of antidiabetic drugs on CEDmean (sd)median [IQR] | 2.12 (0.96)<br>2.00 [1.00, 3.00] | 2.08 (0.96)<br>2.00 [1.00, 3.00] | 0.04 (0.03, 0.05) | 2.08 (0.95)<br>2.00 [1.00, 3.00] | 2.08 (0.96)<br>2.00 [1.00, 3.00] | -0.00 (-0.01, 0.01)<br>- (-, -) |
| Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max | 2.12 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00 | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00 | 0.04 (0.03, 0.05)<br>- (-, -)<br>- (-, -) | 2.08 (0.95)<br>2.00 [1.00, 3.00]<br>1.00, 7.00 | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00 | -0.00 (-0.01, 0.01)<br>- (-, -)<br>- (-, -) |
| Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) | 212 (0.96)<br>200 [1.00, 3.00]<br>1.00, 7.00<br>61,339 (49.3%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,479 (48.3%) | 0.04 (0.03, 0.05)<br>-(-, -)<br>-(-, -)<br>1.0% (0.5%, 1.5%) | 2.08 (0.95)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,467 (48.4%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,388 (48.3%) | -0.00 (-0.01, 0.01)<br>-(-, -)<br>-(-, -)<br>0.1% (-0.4%, 0.7%) |
| Number of antidiabetic drugs on CEDmean (sd)median [IQR]median [IQR]median [IQR]concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) | 212 (0.96)<br>200 (1.00, 3.00)<br>1.00, 7.00<br>61,339 (49.3%)<br>22,397 (18.0%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,479 (48.3%)<br>10,552 (17.3%) | 0.04 (0.03, 0.05)<br>-(-, -)<br>-(-, -)<br>1.0% (0.5%, 1.5%)<br>0.7% (0.4%, 1.1%) | 208 (0.95)<br>200 [1.00, 3.00]<br>1.00, 7.00<br>29,467 (48.4%)<br>10,364 (17.0%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,388 (48.3%)<br>10,510 (17.3%) | -0.00 (-0.01, 0.01)<br>-(-, -)<br>-(-, -)<br>0.1% (-0.4%, 0.7%)<br>-0.2% (-0.7%, 0.2%) |
| Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformir; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) | 2.12 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>61,339 (49.3%)<br>22,397 (18.0%)<br>20,237 (16.3%) | 2.08 (0.96)<br>2.00 (1.00, 3.00)<br>1.00, 7.00<br>29,479 (48.3%)<br>10,552 (17.3%)<br>8,707 (14.3%) | 0.04 (0.03, 0.05)<br>-(-, -)<br>-(-, -)<br>1.0% (0.5%, 1.5%)<br>0.7% (0.4%, 1.1%)<br>2.0% (1.7%, 2.4%) | 2.08 (0.95)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,467 (48.4%)<br>10,364 (17.0%)<br>8,702 (14.3%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,388 (48.3%)<br>10,510 (17.3%)<br>8,694 (14.3%) | -0.00 (-0.01, 0.01)<br>-(-, -)<br>-(-, -)<br>0.1% (-0.4%, 0.7%)<br>-0.2% (-0.7%, 0.2%)<br>0.0% (-0.4%, 0.4%) |
| Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of Sulfonylureas; n (%) | 2.12 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>61,339 (49.3%)<br>22,397 (18.0%)<br>20,237 (16.3%)<br>2,462 (2.0%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,479 (48.3%)<br>10,552 (17.3%)<br>8,707 (14.3%)<br>1.273 (21%) | 0.04 (0.03, 0.05)<br>- (-, -)<br>- (-, -)<br>1.0% (0.5%, 1.5%)<br>0.7% (0.4%, 1.1%)<br>2.0% (1.7%, 2.4%)<br>-0.1% (-0.2%, 0.0%) | 2.08 (0.95)<br>2.00 (1.00, 3.00)<br>1.00, 7.00<br>29,467 (48.4%)<br>10,364 (17.0%)<br>8,702 (14.3%)<br>1,261 (2.1%) | 2.08 (0.96)<br>2.00 (1.00, 3.00)<br>1.00, 7.00<br>29,388 (48.3%)<br>10.510 (17.3%)<br>8.694 (14.3%)<br>1,265 (21%) | -0.00 (-0.01, 0.01)<br>-(-, -)<br>-(-, -)<br>-(-, -)<br>-0.1% (-0.4%, 0.7%)<br>-0.2% (-0.7%, 0.2%)<br>0.0% (-0.4%, 0.4%)<br>-0.0% (-0.2%, 0.2%) |
| Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of DPP-4; n (%) Concomitant use or initiation of SPL-1; n (%) | 2.12 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>61,339 (49.3%)<br>22,397 (18.0%)<br>20,237 (16.3%)<br>2.462 (2.0%)<br>21,296 (17.1%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,479 (48.3%)<br>10,552 (17.3%)<br>8,707 (14.3%)<br>1,273 (21%)<br>10,715 (17.5%) | 0.04 (0.03, 0.05)<br>- (-, -)<br>- (-, -)<br>1.0% (0.5%, 1.5%)<br>0.7% (0.4%, 1.1%)<br>2.0% (1.7%, 2.4%)<br>-0.1% (-0.2%, 0.0%)<br>-0.4% (-0.8%, -0.1%) | 2.08 (0.95)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,467 (48.4%)<br>10,364 (17.0%)<br>8,702 (14.3%)<br>1,261 (21%)<br>10,540 (17.3%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,388 (48.3%)<br>10,510 (17.3%)<br>8.694 (14.3%)<br>1.265 (21%)<br>10,665 (17.5%) | -0.00 (-0.01, 0.01)<br>-(-, -)<br>-(-, -)<br>-0.1% (-0.4%, 0.7%)<br>-0.2% (-0.7%, 0.2%)<br>0.0% (-0.4%, 0.4%)<br>-0.0% (-0.2%, 0.2%)<br>-0.2% (-0.6%, 0.2%) |
| Number of antidiabetic drugs on CEDmean [sd)median [QR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of DPP-4!; n (%) Concomitant use or initiation of SGLT-2!; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) | 2.12 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>61,339 (49.3%)<br>22,397 (18.0%)<br>20,237 (16.3%)<br>2.462 (2.0%)<br>21,296 (17.1%)<br>7,079 (5.7%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,479 (48.3%)<br>10,552 (17.3%)<br>8,707 (14.3%)<br>1,273 (21%)<br>10,715 (17.5%)<br>3,381 (5.5%) | 0.04 (0.03, 0.05)<br>- (-, -)<br>- (-, -)<br>- (-, -)<br>- (-, -)<br>1.0% (0.5%, 1.5%)<br>0.7% (0.4%, 1.1%)<br>2.0% (1.7%, 2.4%)<br>-0.1% (-0.2%, 0.0%)<br>-0.4% (-0.8%, -0.1%)<br>0.2% (-0.1%, 0.4%) | 2.08 (0.95)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,467 (48.4%)<br>10,364 (17.0%)<br>8,702 (14.3%)<br>1,261 (2.1%)<br>10,540 (17.3%)<br>3,342 (5.5%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,388 (48.3%)<br>10,510 (17.3%)<br>8,694 (14.3%)<br>1.265 (21%)<br>10,665 (17.5%)<br>3,369 (5.5%) | -0.00 (-0.01, 0.01) -(-, -) -(-, -) -(-, -) -0.2% (-0.7%, 0.2%) -0.0% (-0.4%, 0.4%) -0.0% (-0.0%, 0.2%) -0.2% (-0.6%, 0.2%) -0.0% (-0.3%, 0.2%) |
| Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max | 212 (0.96)<br>200 [1.00, 3.00]<br>100, 7.00<br>61,339 (49.3%)<br>22,397 (18.0%)<br>20,237 (16.3%)<br>24,62 (2.0%)<br>21,296 (17.1%)<br>7,079 (5.7%)<br>81,498 (65.5%) | 2.08 (0.96)<br>2.00 (1.00, 3.00)<br>1.00, 7.00<br>29,479 (48.3%)<br>10,552 (17.3%)<br>8,707 (14.3%)<br>1,273 (2.1%)<br>10,715 (17.5%)<br>3,381 (5.5%)<br>39,433 (64.5%) | 0.04 (0.03, 0.05)<br>- (-, -)<br>- (-, -)<br>- (-, -)<br>1.0% (0.5%, 1.5%)<br>0.7% (0.4%, 1.1%)<br>2.0% (1.7%, 2.4%)<br>-0.1% (-0.2%, 0.0%)<br>-0.4% (-0.8%, -0.1%)<br>0.2% (-0.1%, 0.4%)<br>0.9% (0.5%, 1.4%) | 208 (0.95)<br>200 [1.00, 3.00]<br>1.00, 7.00<br>29,467 (48.4%)<br>10,364 (17.0%)<br>8,702 (14.3%)<br>1,261 (2.1%)<br>10,540 (17.3%)<br>3,342 (5.5%)<br>39,471 (64.9%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,388 (48.3%)<br>10,510 (17.3%)<br>8,694 (14.3%)<br>1,265 (21%)<br>10,665 (17.5%)<br>3,369 (5.5%)<br>39,301 (64.6%) | -0.00 (-0.01, 0.01)<br>-(-, -)<br>-(-, -)<br>-(-, -)<br>-0.2% (-0.7%, 0.2%)<br>-0.0% (-0.4%, 0.4%)<br>-0.0% (-0.2%, 0.2%)<br>-0.0% (-0.3%, 0.2%)<br>-0.0% (-0.3%, 0.2%)<br>0.3% (-0.3%, 0.8%) |
| Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylures; n (%) Concomitant use or initiation of DPP-4i; n (%) Concomitant use or initiation of SGLT-2i; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Insulins; n (%) Past use of Insulins; n (%) | 2.12 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>61,339 (49.3%)<br>22,397 (18.0%)<br>20,237 (16.3%)<br>2.462 (2.0%)<br>21,296 (17.1%)<br>7,079 (5.7%)<br>81,498 (65.5%)<br>29,354 (23.6%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,479 (48.3%)<br>10,552 (17.3%)<br>8,707 (14.3%)<br>1,273 (21%)<br>10,715 (17.5%)<br>3,381 (5.5%)<br>39,433 (64.5%)<br>13,941 (22.8%) | 0.04 (0.03, 0.05)<br>-(-,-)<br>-(-,-)<br>1.0% (0.5%, 1.5%)<br>0.7% (0.4%, 1.1%)<br>2.0% (1.7%, 2.4%)<br>-0.1% (-0.2%, 0.0%)<br>-0.4% (-0.8%, -0.1%)<br>0.2% (-0.1%, 0.4%)<br>0.9% (0.5%, 1.4%)<br>0.8% (0.4%, 1.2%) | 2.08 (0.95)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,467 (48.4%)<br>10,364 (17.0%)<br>8,702 (14.3%)<br>1,261 (2.1%)<br>10,540 (17.3%)<br>3,342 (5.5%)<br>3,347 (64.9%)<br>13,722 (22.6%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,388 (48.3%)<br>10,510 (17.3%)<br>8,694 (14.3%)<br>1,265 (21%)<br>10,665 (17.5%)<br>3,369 (5.5%)<br>3,369 (6.5%)<br>3,381 (22.8%) | -0.00 (-0.01, 0.01)<br>-(-, -)<br>-(-, -)<br>-0.1% (-0.4%, 0.7%)<br>-0.2% (-0.7%, 0.2%)<br>-0.0% (-0.4%, 0.4%)<br>-0.0% (-0.2%, 0.2%)<br>-0.2% (-0.6%, 0.2%)<br>-0.0% (-0.3%, 0.2%)<br>-0.3% (-0.3%, 0.2%)<br>-0.3% (-0.3%, 0.2%) |
| Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformir; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of SPP-4; n (%) Concomitant use or initiation of DPP-4; n (%) Concomitant use or initiation of SGLT-2; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformir, n (%) Past use of Insulins; n (%) Past use of Sulfonylureas; n (%) | 2.12 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>61,339 (49.3%)<br>22,397 (18.0%)<br>20,237 (16.3%)<br>2.462 (2.0%)<br>21,296 (17.1%)<br>7.079 (5.7%)<br>81,498 (65.5%)<br>29,354 (23.6%)<br>28,787 (23.1%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,479 (48.3%)<br>10.552 (17.3%)<br>8,707 (14.3%)<br>1.273 (21%)<br>10,715 (17.5%)<br>3,381 (5.5%)<br>39,433 (64.5%)<br>13,941 (22.8%)<br>12,606 (20.6%) | 0.04 (0.03, 0.05)<br>- (-, -)<br>- (-, -)<br>1.0% (0.5%, 1.5%)<br>0.7% (0.4%, 1.1%)<br>2.0% (1.7%, 2.4%)<br>-0.1% (-0.2%, 0.0%)<br>-0.4% (-0.8%, -0.1%)<br>0.2% (-0.1%, 0.4%)<br>0.9% (0.5%, 1.4%)<br>0.8% (0.4%, 1.2%)<br>2.5% (2.1%, 2.9%) | 2.08 (0.95)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,467 (48.4%)<br>10,364 (17.0%)<br>8,702 (14.3%)<br>1,261 (21%)<br>10,540 (17.3%)<br>3,342 (5.5%)<br>39,471 (64.9%)<br>13,722 (22.6%)<br>12,605 (20.7%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,388 (48.3%)<br>10,510 (17.3%)<br>8.694 (14.3%)<br>1.265 (21%)<br>10,665 (17.5%)<br>3,369 (5.5%)<br>39,301 (64.6%)<br>13,881 (22.8%)<br>12,581 (20.7%) | -0.00 (-0.01, 0.01) -(-, -) -(-, -) -(-, -) -0.1% (-0.4%, 0.7%) -0.2% (-0.7%, 0.2%) -0.0% (-0.4%, 0.4%) -0.0% (-0.2%, 0.2%) -0.2% (-0.6%, 0.2%) -0.0% (-0.3%, 0.2%) -0.0% (-0.3%, 0.2%) -0.0% (-0.3%, 0.8%) -0.3% (-0.7%, 0.2%) -0.3% (-0.7%, 0.2%) |
| Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of DPP-41; n (%) Concomitant use or initiation of SoLT-2; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformin; n (%) Past use of Insulins; n (%) Past use of Sulfonylureas; n (%) Past use of DPP-41; n (%) | 2.12 (0.96) 2.00 [1.00, 3.00] 1.00, 7.00 61,339 (49.3%) 22,397 (16.3%) 2,462 (2.0%) 21,296 (17.1%) 7,079 (5.7%) 81,498 (65.5%) 29,354 (23.6%) 28,787 (23.1%) 4,186 (3.4%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,479 (48.3%)<br>10,552 (17.3%)<br>8,707 (14.3%)<br>1,273 (2.1%)<br>10,715 (17.5%)<br>3,381 (5.5%)<br>39,433 (64.5%)<br>13,941 (22.8%)<br>12,606 (20.6%)<br>2,226 (3.6%) | 0.04 (0.03, 0.05)<br>- (-, -)<br>- (-, -)<br>- (-, -)<br>- (-, -)<br>1.0% (0.5%, 1.5%)<br>0.7% (0.4%, 1.1%)<br>2.0% (1.7%, 2.4%)<br>-0.1% (-0.2%, 0.01%)<br>0.4% (-0.8%, -0.1%)<br>0.2% (-0.1%, 0.4%)<br>0.9% (0.5%, 1.4%)<br>0.8% (0.4%, 1.2%)<br>2.5% (2.1%, 2.9%)<br>-0.3% (-0.5%, -0.1%) | 2.08 (0.95)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,467 (48.4%)<br>10,364 (17.0%)<br>8,702 (14.3%)<br>1,261 (2.1%)<br>10,540 (17.3%)<br>3,342 (5.5%)<br>39,471 (64.9%)<br>13,722 (22.6%)<br>12,605 (20.7%)<br>2,230 (3.7%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,388 (48.3%)<br>10,510 (17.3%)<br>8,694 (14.3%)<br>11,265 (21%)<br>10,665 (17.5%)<br>3,369 (5.5%)<br>39,301 (64.6%)<br>13,881 (22.8%)<br>12,581 (20.7%)<br>2,209 (3.6%) | -0.00 (-0.01, 0.01) -(-, -) -(-, -) -(-, -) -(-, -) -(-, -) -0.2% (-0.7%, 0.2%) -0.0% (-0.4%, 0.4%) -0.0% (-0.2%, 0.2%) -0.2% (-0.6%, 0.2%) -0.0% (-0.3%, 0.2%) -0.3% (-0.3%, 0.2%) -0.3% (-0.3%, 0.2%) -0.0% (-0.4%, 0.2%) -0.0% (-0.4%, 0.2%) -0.0% (-0.4%, 0.2%) |
| Number of antidiabetic drugs on CEDmean [sd]median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of DPP-4i; n (%) Concomitant use or initiation of SGLT-2i; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformin; n (%) Past use of Insulins; n (%) Past use of Sulfonylureas; n (%) Past use of SURFON, in (%) | 212 (0.96) 200 [1.00, 3.00] 1.00, 7.00 61,339 (49.3%) 22,397 (16.3%) 20,237 (16.3%) 2.462 (2.0%) 21,296 (17.1%) 7,079 (5.7%) 31,498 (65.5%) 29,354 (23.6%) 28,787 (23.1%) 4,186 (3.4%) 29,247 (23.5%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,479 (48.3%)<br>10,552 (17.3%)<br>8,707 (14.3%)<br>1,273 (2.1%)<br>10,715 (17.5%)<br>3,381 (5.5%)<br>39,433 (64.5%)<br>13,941 (22.8%)<br>12,606 (20.6%)<br>2,226 (3.6%)<br>14,886 (24.4%) | 0.04 (0.03, 0.05)<br>-(-,-)<br>-(-,-)<br>1.0% (0.5%, 1.5%)<br>0.7% (0.4%, 1.1%)<br>2.0% (1.7%, 2.4%)<br>-0.1% (-0.2%, 0.0%)<br>-0.4% (-0.8%, -0.1%)<br>0.2% (-0.1%, 0.4%)<br>0.9% (0.5%, 1.4%)<br>0.8% (0.4%, 1.2%)<br>2.5% (2.1%, 2.9%)<br>-0.3% (-0.5%, -0.1%)<br>-0.9% (-0.5%, -0.1%) | 2.08 (0.95)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,467 (48.4%)<br>10,364 (17.0%)<br>8,702 (14.3%)<br>1,261 (2.1%)<br>10,540 (17.3%)<br>3,342 (5.5%)<br>39,471 (64.9%)<br>13,722 (22.6%)<br>12,605 (20.7%)<br>2,230 (3.7%)<br>14,735 (24.2%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,388 (48.3%)<br>10,510 (17.3%)<br>8.694 (14.3%)<br>1,265 (21%)<br>10,665 (17.5%)<br>33,369 (5.5%)<br>39,301 (64.6%)<br>13,881 (22.8%)<br>12,581 (20.7%)<br>2,209 (3.6%)<br>14,812 (24.3%) | -0.00 (-0.01, 0.01) -(-, -) -(-, -) -(-, -) -(-, -) -(-, -) -0.2% (-0.7%, 0.2%) -0.0% (-0.4%, 0.4%) -0.0% (-0.2%, 0.2%) -0.0% (-0.3%, 0.2%) -0.3% (-0.3%, 0.2%) -0.3% (-0.3%, 0.8%) -0.3% (-0.7%, 0.2%) -0.0% (-0.2%, 0.2%) -0.0% (-0.2%, 0.2%) -0.0% (-0.2%, 0.2%) |
| Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylures; n (%) Concomitant use or initiation of DPP-4i; n (%) Concomitant use or initiation of DPP-4i; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformin; n (%) Past use of Insulins; n (%) Past use of Sulfonylureas; n (%) Past use of DPP-4i; n (%) Past use of DPP-4i; n (%) Past use of SDP-4i; n (%) Past use of SDP-4i; n (%) Past use of Any other glucose-lowering drugs; n (%) | 2.12 (0.96) 2.00 [1.00, 3.00] 1.00, 7.00 61,339 (49.3%) 22,397 (18.0%) 20,237 (16.3%) 2.462 (2.0%) 21,296 (17.1%) 7.079 (5.7%) 31.498 (65.5%) 29,354 (23.6%) 28,787 (23.1%) 4,186 (3.4%) 29,247 (23.5%) 9,773 (7.9%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,479 (48.3%)<br>10,552 (17.3%)<br>8,707 (14.3%)<br>1,273 (21%)<br>10,715 (17.5%)<br>3,381 (5.5%)<br>39,433 (64.5%)<br>13,941 (22.8%)<br>12,606 (20.6%)<br>2,226 (3.6%)<br>4,756 (7.8%) | 0.04 (0.03, 0.05) -(-,-) -(-,-) 1.0% (0.5%, 1.5%) 0.7% (0.4%, 1.1%) 2.0% (1.7%, 2.4%) -0.1% (-0.2%, 0.0%) -0.4% (-0.8%, -0.1%) 0.2% (-0.1%, 0.4%) 0.9% (0.5%, 1.4%) 0.8% (0.4%, 1.2%) 2.5% (21%, 2.9%) -0.3% (-0.5%, -0.1%) 0.9% (-1.3%, -0.5%) 0.1% (-0.2%, 0.3%) | 2.08 (0.95)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,467 (48.4%)<br>10,364 (17.0%)<br>8,702 (14.3%)<br>1.261 (21%)<br>10,540 (17.3%)<br>3,342 (5.5%)<br>33,471 (64.9%)<br>13,722 (22.6%)<br>12,605 (20.7%)<br>2,230 (3.7%)<br>14,735 (24.2%)<br>4,746 (7.8%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,388 (48.3%)<br>10,510 (17.3%)<br>8,694 (14.3%)<br>1,255 (21%)<br>10,665 (17.5%)<br>3,369 (5.5%)<br>33,301 (64.6%)<br>13,881 (22.8%)<br>12,581 (20.7%)<br>2,209 (3.6%)<br>14,812 (24.3%)<br>4,739 (7.8%) | -0.00 (-0.01, 0.01) -(-, -) -(-, -) -(-, -) -0.2% (-0.7%, 0.2%) -0.2% (-0.7%, 0.2%) -0.0% (-0.4%, 0.4%) -0.0% (-0.2%, 0.2%) -0.2% (-0.6%, 0.2%) -0.3% (-0.3%, 0.2%) -0.3% (-0.3%, 0.5%) -0.3% (-0.3%, 0.5%) -0.3% (-0.0.7%, 0.2%) -0.0% (-0.0.7%, 0.2%) -0.0% (-0.0.7%, 0.2%) -0.0% (-0.0.7%, 0.2%) |
| Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformir; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of SPP-4; n (%) Concomitant use or initiation of DPP-4; n (%) Concomitant use or initiation of SGLT-2; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformin; n (%) Past use of Sulfonylureas; n (%) Past use of SPP-4; n (%) Past use of SPP-4; n (%) Past use of SGLT-2; n (%) Past use of SGT-2; n (%) Past use of SGRT-2; n (%) | 212 (0.96) 200 [1.00, 3.00] 1.00, 7.00 61,339 (49.3%) 22,397 (18.0%) 20,237 (16.3%) 24,62 (2.0%) 21,296 (17.1%) 7.079 (5.7%) 81,498 (65.5%) 29,354 (23.6%) 28,787 (23.1%) 4,186 (3.4%) 29,247 (23.5%) 9,737 (7.9%) 90,662 (72.8%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,479 (48.3%)<br>10.552 (17.3%)<br>8,707 (14.3%)<br>1.273 (21%)<br>10,715 (17.5%)<br>3,381 (5.5%)<br>39,433 (64.5%)<br>13,941 (22.8%)<br>12,606 (20.6%)<br>2,226 (3.6%)<br>14,886 (24.4%)<br>4,756 (7.8%)<br>43,860 (71.8%) | 0.04 (0.03, 0.05) -(-,-) -(-,-) 1.0% (0.5%, 1.5%) 0.7% (0.4%, 1.1%) 2.0% (1.7%, 2.4%) -0.1% (-0.2%, 0.0%) -0.4% (-0.8%, -0.1%) 0.2% (-0.1%, 0.4%) 0.9% (0.5%, 1.4%) 0.9% (0.5%, 1.4%) 0.5% (2.1%, 2.9%) -0.3% (-0.5%, -0.1%) -0.3% (-0.5%, -0.1%) 0.9% (1.3%, -0.5%) 0.1% (-0.2%, 0.3%) | 2.08 (0.95)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,467 (48.4%)<br>10,364 (17.0%)<br>8,702 (14.3%)<br>1,261 (21%)<br>10,540 (17.3%)<br>3,342 (5.5%)<br>39,471 (64.9%)<br>13,722 (22.6%)<br>12,605 (20.7%)<br>2,230 (3.7%)<br>14,735 (24.2%)<br>4,746 (7.8%)<br>43,638 (71.7%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,388 (48.3%)<br>10,510 (17.3%)<br>8.694 (14.3%)<br>1.265 (21%)<br>10,665 (17.5%)<br>33.69 (5.5%)<br>39,301 (64.6%)<br>13,881 (22.8%)<br>12,581 (20.7%)<br>2,209 (3.6%)<br>14,812 (24.3%)<br>4,739 (7.8%)<br>43,704 (71.8%) | -0.00 (-0.01, 0.01) -(-, -) -( |
| Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformir; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of SPP-4i; n (%) Concomitant use or initiation of SPP-4i; n (%) Concomitant use or initiation of SGLT-2j; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformir; n (%) Past use of Insulins; n (%) Past use of Sulfonylureas; n (%) Past use of Sulfonylureas; n (%) Past use of SGLT-2j; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ARNI; n (%) ARNI; n (%) | 2.12 (0.96) 2.00 [1.00, 3.00] 1.00, 7.00 61,339 (49.3%) 22,397 (18.0%) 20,237 (16.3%) 2.462 (2.0%) 21,296 (17.1%) 7.079 (5.7%) 81,498 (65.5%) 29,354 (23.6%) 28,787 (23.1%) 4,186 (3.4%) 29,247 (23.5%) 9,773 (7.9%) 9,0662 (72.8%) 2,404 (1.9%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,479 (48.3%)<br>10,552 (17.3%)<br>8,707 (14.3%)<br>1,273 (2.1%)<br>10,715 (17.5%)<br>3,381 (5.5%)<br>39,433 (64.5%)<br>12,606 (20.6%)<br>2,226 (3.6%)<br>14,886 (24.4%)<br>4,756 (7.8%)<br>4,860 (71.8%)<br>1,058 (1.7%) | 0.04 (0.03, 0.05) -(-, -) -(-, -) -(-, -) -(-, -) 1.0% (0.5%, 1.5%) 0.7% (0.4%, 1.1%) 2.0% (1.7%, 2.4%) -0.1% (-0.2%, 0.0%) 0.4% (-0.2%, 0.0%) 0.2% (-0.1%, 0.4%) 0.2% (0.1%, 1.4%) 0.2% (0.4%, 1.2%) 2.5% (2.1%, 2.9%) -0.3% (-0.5%, -0.1%) 0.9% (1.3%, -0.5%) 0.1% (-0.5%, -0.1%) | 2.08 (0.95)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,467 (48.4%)<br>10,364 (17.0%)<br>8,702 (14.3%)<br>1,261 (21%)<br>10,540 (17.3%)<br>3,342 (5.5%)<br>39,471 (64.9%)<br>12,605 (20.7%)<br>2,230 (3.7%)<br>14,735 (24.2%)<br>4,746 (7.8%)<br>4,3638 (71.7%)<br>1,068 (1.8%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,388 (48.3%)<br>10,510 (17.3%)<br>8.694 (14.3%)<br>11,265 (21%)<br>10,665 (17.5%)<br>3,369 (5.5%)<br>39,301 (64.6%)<br>12,581 (20.7%)<br>2,209 (3.6%)<br>14,812 (24.3%)<br>4,739 (7.8%)<br>4,739 (7.8%)<br>1,058 (1.7%) | -0.00 (-0.01, 0.01) -(-, -) -( |
| Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of SGLT-2i; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Insulins; n (%) Past use of Insulins; n (%) Past use of SelT-2i; n (%) Past use of DPP-4i; n (%) Past use of Any other glucose-lowering drugs; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ARNI; n (%) Thiazides; n (%) Thiazides; n (%) | 212 (0.96) 210 [1.00, 3.00] 100, 7.00 61,339 (49.3%) 22,397 (8.0%) 22,397 (16.3%) 24,62 (2.0%) 21,296 (17.1%) 7,079 (5.7%) 81,498 (65.5%) 29,354 (23.6%) 28,787 (23.1%) 41,86 (3.4%) 29,247 (23.5%) 9,773 (7.9%) 90,662 (72.8%) 2404 (1.9%) 43,619 (35.0%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,479 (48.3%)<br>10,552 (17.3%)<br>8,707 (14.3%)<br>1,273 (2.1%)<br>10,715 (17.5%)<br>3,381 (5.5%)<br>39,433 (64.5%)<br>13,941 (22.8%)<br>12,606 (20.6%)<br>2,226 (3.6%)<br>14,886 (24.4%)<br>4,756 (7.8%)<br>43,860 (71.8%)<br>1,058 (17.9%)<br>21,633 (35.4%) | 0.04 (0.03, 0.05) -(-,-) -(-,-) 1.0% (0.5%, 1.5%) 0.7% (0.4%, 1.1%) 2.0% (1.7%, 2.4%) -0.16 (-0.2%, 0.0%) -0.4% (-0.8%, -0.1%) 0.2% (-0.1%, 0.4%) 0.9% (0.5%, 1.4%) 0.8% (0.4%, 1.2%) 2.5% (2.1%, 2.9%) -0.3% (-0.5%, -0.1%) 0.9% (0.5%, 1.5%) 0.1% (-0.2%, 0.3%) 1.0% (0.6%, 1.5%) 0.2% (0.6%, 1.5%) | 2.08 (0.95)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,467 (48.4%)<br>10.364 (17.0%)<br>8.702 (14.3%)<br>1.261 (21%)<br>10.540 (17.3%)<br>3.342 (5.5%)<br>33,471 (64.9%)<br>13,722 (22.6%)<br>12,605 (20.7%)<br>2.230 (3.7%)<br>14,735 (24.2%)<br>4,746 (7.8%)<br>43,638 (71.7%)<br>1.068 (1.8%)<br>21,701 (35.7%) | 2.08 (0.96)<br>2.00 (1.00, 3.00)<br>1.00, 7.00<br>29,388 (48.3%)<br>10.510 (17.3%)<br>8.694 (14.3%)<br>1,265 (21%)<br>10,665 (17.5%)<br>3,369 (5.5%)<br>33,391 (64.6%)<br>13,881 (22.8%)<br>12,581 (20.7%)<br>22,209 (3.6%)<br>14,812 (24.3%)<br>4,739 (7.8%)<br>1,058 (1.7%)<br>21,551 (35.4%) | -0.00 (-0.01, 0.01) -(-, -) -(-, -) -(-, -) -(-, -) -(-, -) -(-, -) -0.2% (-0.7%, 0.2%) -0.2% (-0.7%, 0.2%) -0.0% (-0.2%, 0.2%) -0.2% (-0.6%, 0.2%) -0.0% (-0.3%, 0.2%) -0.0% (-0.3%, 0.2%) -0.0% (-0.3%, 0.2%) -0.0% (-0.3%, 0.2%) -0.0% (-0.3%, 0.2%) -0.0% (-0.4%, 0.5%) -0.0% (-0.2%, 0.2%) -0.1% (-0.6%, 0.4%) -0.0% (-0.3%, 0.3%) -0.1% (-0.6%, 0.4%) -0.0% (-0.3%, 0.3%) -0.1% (-0.6%, 0.4%) -0.0% (-0.3%, 0.3%) |
| Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of SP-4; n (%) Concomitant use or initiation of SP-4; n (%) Concomitant use or initiation of SP-4; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformin; n (%) Past use of Self-12; n (%) Past use of Self-12; n (%) Past use of Self-12; n (%) Past use of Self-12; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-13/ARB's; n (%) ARN; n (%) Thiazides; n (%) Beta-blockers; n (%) Beta-blockers; n (%) | 212 (0.96) 200 [1.00, 3.00] 1.00, 7.00 61,339 (49.3%) 22,397 (18.0%) 20,237 (16.3%) 2,462 (2.0%) 21,296 (17.1%) 7,079 (5.7%) 31,498 (65.5%) 29,354 (23.6%) 28,787 (23.1%) 4,186 (3.4%) 29,247 (23.5%) 9,773 (7.9%) 90,662 (72.8%) 2,404 (1.9%) 4,3619 (35.0%) 53,555 (43.0%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,479 (48.3%)<br>10,552 (17.3%)<br>8,707 (14.3%)<br>1,273 (21%)<br>10,715 (17.5%)<br>3,381 (5.5%)<br>39,433 (64.5%)<br>13,941 (22.8%)<br>12,606 (20.6%)<br>2,226 (3.6%)<br>14,886 (24.4%)<br>4,756 (7.8%)<br>43,860 (71.8%)<br>10,58 (1.7%)<br>21,633 (35.4%)<br>24,449 (40.0%) | 0.04 (0.03, 0.05) -(-,-) -(-,-) 1.0% (0.5%, 1.5%) 0.7% (0.4%, 1.1%) 2.0% (1.7%, 2.4%) -0.1% (-0.2%, 0.0%) -0.4% (-0.9%, -0.1%) 0.2% (-0.1%, 0.4%) 0.9% (0.5%, 1.4%) 0.8% (0.5%, 1.4%) 0.8% (0.4%, 1.2%) 2.5% (2.1%, 2.9%) -0.3% (-0.5%, -0.1%) 0.09% (1.3%, 0.5%) 0.1% (-0.2%, 0.3%) 0.1% (-0.2%, 0.3%) 0.2% (0.5%, 1.5%) 0.2% (0.5%, 1.5%) 0.2% (0.5%, 1.5%) | 2.08 (0.95) 2.00 [1.00, 3.00] 1.00, 7.00 29,467 (48.4%) 10,364 (17.0%) 8.702 (14.3%) 1.261 (21%) 10,540 (17.3%) 3,342 (5.5%) 33,471 (64.9%) 13,722 (22.6%) 12,605 (20.7%) 2.230 (3.7%) 14,735 (24.2%) 4,746 (7.8%) 43,638 (71.7%) 1.068 (1.8%) 2,1701 (35.7%) 24,381 (40.1%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,388 (48.3%)<br>10,510 (17.3%)<br>8.694 (14.3%)<br>1,255 (21%)<br>10,665 (17.5%)<br>3,369 (5.5%)<br>3,369 (5.5%)<br>13,881 (22.8%)<br>12,581 (20.7%)<br>2.209 (3.6%)<br>14,812 (24.3%)<br>4,739 (7.8%)<br>4,739 (7.8%)<br>1,058 (1.7%)<br>2,515 (135.4%)<br>24,395 (40.1%) | -0.00 (-0.01, 0.01) -(-, -) -( |
| Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformir; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of SP-4; n (%) Concomitant use or initiation of DPP-4; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformir, n (%) Past use of Sulfonylureas; n (%) Past use of SPP-4; n (%) Past use of SPP-4; n (%) Past use of SPP-4; n (%) Past use of SPP-4; n (%) ACE-is/ARB's; n (%) ACE-is/ARB's; n (%) ARN; n (%) Thiazides; n (%) Beta blockers; n (%) Calcium channel blockers; n (%) | 212 (0.96) 200 [1.00, 3.00] 1.00, 7.00 61.339 (49.3%) 22.397 (18.0%) 20.237 (16.3%) 2.462 (2.0%) 21.296 (17.1%) 7.079 (5.7%) 81.498 (65.5%) 29.354 (23.6%) 28.787 (23.1%) 4,186 (3.4%) 29.247 (23.5%) 9,773 (7.9%) 90.662 (72.8%) 2404 (1.9%) 43.619 (35.0%) 53.555 (43.0%) 41.983 (33.7%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,479 (48.3%)<br>10.552 (17.3%)<br>8,707 (14.3%)<br>1.273 (21%)<br>10,715 (17.5%)<br>3,381 (5.5%)<br>39,433 (64.5%)<br>13,941 (22.8%)<br>12,606 (20.6%)<br>2,226 (3.6%)<br>14,886 (24.4%)<br>4,756 (7.8%)<br>43,860 (71.8%)<br>1,058 (1.7%)<br>21,633 (35.4%)<br>24,449 (40.0%)<br>19,388 (31.7%) | 0.04 (0.03, 0.05) -(-,-) -(-,-) 1.0% (0.5%, 1.5%) 0.7% (0.4%, 1.1%) 2.0% (1.7%, 2.4%) -0.1% (-0.2%, 0.0%) -0.4% (-0.8%, -0.1%) 0.2% (-0.1%, 0.4%) 0.9% (0.5%, 1.4%) 0.9% (0.5%, 1.4%) 0.9% (0.5%, 1.4%) 0.9% (0.5%, 0.1%) -0.3% (-0.5%, 0.1%) -0.3% (-0.5%, 0.1%) -0.9% (1.3%, -0.5%) 0.1% (-0.2%, 0.3%) 1.0% (0.6%, 1.5%) 0.2% (0.1%, 0.3%) -0.4% (-0.8%, 0.1%) 3.0% (2.5%, 3.5%) | 2.08 (0.95) 2.00 [1.00, 3.00] 1.00, 7.00 29.467 (48.4%) 10.364 (17.0%) 8,702 (14.3%) 1,261 (21%) 10,540 (17.3%) 3,342 (5.5%) 39.471 (64.9%) 13,722 (22.6%) 12,605 (20.7%) 2,230 (3.7%) 14,735 (24.2%) 4,746 (7.8%) 43,638 (71.7%) 1,068 (1.8%) 21,701 (35.7%) 24,381 (40.1%) 19,378 (31.8%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,388 (48.3%)<br>10,510 (17.3%)<br>8.694 (14.3%)<br>1.265 (21%)<br>10,665 (17.5%)<br>3.369 (5.5%)<br>39,301 (64.6%)<br>13,881 (22.8%)<br>12,581 (20.7%)<br>2.209 (3.6%)<br>14,812 (24.3%)<br>4,739 (7.8%)<br>43,704 (71.8%)<br>1.058 (1.7%)<br>21,551 (35.4%)<br>24,395 (40.1%)<br>19,342 (31.8%) | -0.00 (-0.01, 0.01) -(-, -) -( |
| Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformir; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of DPP-4i; n (%) Concomitant use or initiation of SGLT-2i; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformir; n (%) Past use of Insulins; n (%) Past use of Sulfonylureas; n (%) Past use of Sulfonylureas; n (%) Past use of SGLT-2i; n (%) Past use of Any other glucose-lowering drugs; n (%) ARNI; n (%) Thiazides; n (%) Beta-blockers; n (%) Calcium channel blockers; n (%) Digoxin / Digitoxin; n (%) | 212 (0.96) 200 [1.00, 3.00] 1.00, 7.00 61,339 (49.3%) 22,397 (18.0%) 20,237 (16.3%) 2,462 (2.0%) 21,296 (17.1%) 7,079 (5.7%) 81,498 (65.5%) 29,354 (23.6%) 28,787 (23.1%) 4,186 (3.4%) 29,247 (23.5%) 9,773 (7.9%) 90,662 (72.8%) 2,404 (1.9%) 43,619 (35.0%) 53,555 (43.0%) 41,983 (33.7%) 698 (0.6%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,479 (48.3%)<br>10,552 (17.3%)<br>8,707 (14.3%)<br>1.273 (2.1%)<br>10,715 (17.5%)<br>3,381 (5.5%)<br>39,433 (64.5%)<br>12,606 (20.6%)<br>2,226 (3.6%)<br>14,886 (24.4%)<br>4,756 (7.8%)<br>43,860 (71.8%)<br>1,058 (1.7%)<br>24,449 (40.0%)<br>19,388 (31.7%)<br>303 (0.5%) | 0.04 (0.03, 0.05) -(-,-) -(-,-) -(-,-) 1.0% (0.5%, 1.5%) 0.7% (0.4%, 1.15%) 2.0% (1.7%, 2.4%) -0.1% (-0.2%, 0.0%) -0.4% (-0.8%, -0.1%) 0.2% (-0.1%, 0.4%) 0.9% (0.5%, 1.4%) 0.9% (0.5%, 1.4%) 0.9% (0.5%, 1.4%) -0.9% (0.3%, -0.1%) -0.9% (1.3%, -0.5%) 0.1% (-0.5%, -0.1%) -0.9% (1.3%, -0.5%) 0.1% (-0.5%, -0.1%) -0.9% (1.3%, -0.5%) 0.2% (0.1%, 0.3%) -0.4% (-0.8%, 0.1%) 3.0% (2.5%, 3.5%) 2.0% (1.5%, 2.4%) 0.1% (-0.0%, 0.1%) | 2.08 (0.95) 2.00 [1.00, 3.00] 1.00, 7.00 29.467 (48.4%) 10,364 (17.0%) 8,702 (14.3%) 1.261 (21%) 10,540 (17.3%) 3,342 (5.5%) 39.471 (64.9%) 13,722 (22.6%) 12,605 (20.7%) 2,230 (3.7%) 14,735 (24.2%) 4,746 (7.8%) 4,3638 (71.7%) 1.068 (1.8%) 21,701 (35.7%) 24,381 (40.1%) 19,378 (31.8%) 300 (0.5%) | 2.08 (0.96) 2.00 [1.00, 3.00] 1.00, 7.00 29,388 (48.3%) 10,510 (17.3%) 8.694 (14.3%) 1.265 (21%) 10,665 (17.5%) 3,369 (5.5%) 39,301 (64.6%) 13,881 (22.8%) 12,581 (20.7%) 2.209 (3.6%) 14,812 (24.3%) 4,739 (7.8%) 4,739 (7.8%) 1,058 (1.7%) 21,551 (35.4%) 24,395 (40.1%) 19,342 (31.8%) 302 (0.5%) | -0.00 (-0.01, 0.01) -(-, -) -( |
| Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of SPP-4i; n (%) Concomitant use or initiation of SPP-4i; n (%) Concomitant use or initiation of SPP-4i; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Insulins; n (%) Past use of Insulins; n (%) Past use of Sulfonylureas; n (%) Past use of Sulfonylureas; n (%) Past use of SPP-4i; n (% | 212 (0.96) 210 [1.00, 3.00] 1.00, 7.00 61,339 (49.3%) 22,397 (18.0%) 20,237 (16.3%) 24.62 (2.0%) 21,296 (17.1%) 7,079 (5.7%) 81.498 (65.5%) 29,354 (23.6%) 28,787 (23.1%) 4,186 (3.4%) 29,247 (23.5%) 9,773 (7.9%) 90,662 (72.8%) 24.04 (1.9%) 43.619 (35.0%) 53,555 (43.0%) 41,983 (33.7%) 698 (0.6%) 23,870 (19.2%) | 2.08 (0.96) 2.00 [1.00, 3.00] 1.00, 7.00 29,479 (48.3%) 10.552 (17.3%) 8.707 (14.3%) 1.273 (21%) 10.715 (17.5%) 3.381 (5.5%) 39,433 (64.5%) 13,941 (22.8%) 12.606 (20.6%) 2.226 (3.6%) 43,860 (71.8%) 4,756 (7.8%) 43,860 (71.8%) 1,058 (1.7%) 21,633 (35.4%) 24,449 (40.0%) 19,388 (31.7%) 303 (0.5%) 10,613 (17.4%) | 0.04 (0.03, 0.05) -(-,-) -(-,-) 1.0% (0.5%, 1.5%) 0.7% (0.4%, 1.1%) 2.0% (1.7%, 2.4%) -0.1% (-0.2%, 0.0%) -0.4% (-0.8%, -0.1%) 0.2% (-0.1%, 0.4%) 0.2% (-0.5%, 1.4%) 0.8% (0.4%, 1.2%) 2.5% (2.1%, 2.9%) -0.3% (-0.5%, -0.1%) -0.3% (-0.5%, -0.1%) 0.0% (0.5%, 1.4%) 0.8% (0.4%, 1.2%) 2.5% (2.1%, 2.9%) -0.3% (-0.5%, 0.1%) -0.3% (-0.5%, 0.1%) 3.0% (2.5%, 3.5%) 0.4% (-0.8%, 0.1%) 3.0% (2.5%, 3.5%) 2.0% (1.5%, 2.4%) 0.1% (-0.9%, 0.1%) 3.0% (2.5%, 3.5%) | 2.08 (0.95) 2.00 [1.00, 3.00] 1.00, 7.00 29,467 (48.4%) 10.364 (17.0%) 8.702 (14.3%) 1.261 (2.1%) 10,540 (17.3%) 3.342 (5.5%) 3.342 (5.5%) 3.342 (5.5%) 12,605 (20.7%) 12,605 (20.7%) 12,605 (20.7%) 14,735 (24.2%) 4,746 (7.8%) 43,638 (71.7%) 10,68 (1.8%) 21,701 (35.7%) 24,381 (40.1%) 19,378 (31.8%) 19,378 (31.8%) 10,709 (17.6%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,388 (48.3%)<br>10,510 (17.3%)<br>8.694 (14.3%)<br>1,265 (21%)<br>10,665 (17.5%)<br>3,369 (5.5%)<br>33,391 (64.6%)<br>13,881 (22.8%)<br>12,581 (20.7%)<br>2,209 (3.6%)<br>14,812 (24.3%)<br>4,739 (7.8%)<br>4,739 (7.8%)<br>21,551 (35.4%)<br>24,395 (40.1%)<br>19,342 (31.8%)<br>302 (0.5%)<br>10,598 (17.4%) | -0.00 (-0.01, 0.01) -(-, -) -(-, -) -(-, -) -(-, -) -(-, -) -(-, -) -0.2% (-0.7%, 0.2%) -0.2% (-0.7%, 0.2%) -0.0% (-0.2%, 0.2%) -0.0% (-0.2%, 0.2%) -0.0% (-0.3%, 0.2%) -0.3% (-0.3%, 0.2%) -0.0% (-0.2%, 0.2%) -0.1% (-0.6%, 0.4%) -0.0% (-0.3%, 0.3%) -0.1% (-0.6%, 0.4%) -0.0% (-0.3%, 0.3%) -0.0% (-0.3%, 0.5%) -0.0% (-0.3%, 0.5%) -0.0% (-0.5%, 0.5%) -0.0% (-0.5%, 0.5%) |
| Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformir; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of DPP-4i; n (%) Concomitant use or initiation of SGLT-2i; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformir; n (%) Past use of Insulins; n (%) Past use of Sulfonylureas; n (%) Past use of Sulfonylureas; n (%) Past use of SGLT-2i; n (%) Past use of Any other glucose-lowering drugs; n (%) ARNI; n (%) Thiazides; n (%) Beta-blockers; n (%) Calcium channel blockers; n (%) Digoxin / Digitoxin; n (%) | 212 (0.96) 200 [1.00, 3.00] 1.00, 7.00 61,339 (49.3%) 22,397 (18.0%) 20,237 (16.3%) 2,462 (2.0%) 21,296 (17.1%) 7,079 (5.7%) 81,498 (65.5%) 29,354 (23.6%) 28,787 (23.1%) 4,186 (3.4%) 29,247 (23.5%) 9,773 (7.9%) 90,662 (72.8%) 2,404 (1.9%) 43,619 (35.0%) 53,555 (43.0%) 41,983 (33.7%) 698 (0.6%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,479 (48.3%)<br>10,552 (17.3%)<br>8,707 (14.3%)<br>1.273 (2.1%)<br>10,715 (17.5%)<br>3,381 (5.5%)<br>39,433 (64.5%)<br>12,606 (20.6%)<br>2,226 (3.6%)<br>14,886 (24.4%)<br>4,756 (7.8%)<br>43,860 (71.8%)<br>1,058 (1.7%)<br>24,449 (40.0%)<br>19,388 (31.7%)<br>303 (0.5%) | 0.04 (0.03, 0.05) -(-, -) -(-, -) -(-, -) 1.0% (0.5%, 1.5%) 0.7% (0.4%, 1.15%) 2.0% (1.7%, 2.4%) -0.1% (-0.2%, 0.0%) -0.4% (-0.8%, -0.1%) 0.2% (-0.1%, 0.4%) 0.9% (0.5%, 1.4%) 0.9% (0.5%, 1.4%) 0.9% (0.5%, 1.4%) -0.9% (0.3%, -0.1%) -0.9% (1.3%, -0.5%) 0.1% (-0.5%, -0.1%) -0.9% (1.3%, -0.5%) 0.1% (-0.5%, -0.1%) -0.9% (1.3%, -0.5%) 0.2% (0.1%, 0.3%) -0.4% (-0.8%, 0.1%) 3.0% (2.5%, 3.5%) 2.0% (1.5%, 2.4%) 0.1% (-0.0%, 0.1%) | 2.08 (0.95) 2.00 [1.00, 3.00] 1.00, 7.00 29.467 (48.4%) 10,364 (17.0%) 8,702 (14.3%) 1.261 (21%) 10,540 (17.3%) 3,342 (5.5%) 39.471 (64.9%) 13,722 (22.6%) 12,605 (20.7%) 2,230 (3.7%) 14,735 (24.2%) 4,746 (7.8%) 4,3638 (71.7%) 1.068 (1.8%) 21,701 (35.7%) 24,381 (40.1%) 19,378 (31.8%) 300 (0.5%) | 2.08 (0.96) 2.00 [1.00, 3.00] 1.00, 7.00 29,388 (48.3%) 10,510 (17.3%) 8.694 (14.3%) 1.265 (21%) 10,665 (17.5%) 3,369 (5.5%) 39,301 (64.6%) 13,881 (22.8%) 12,581 (20.7%) 2.209 (3.6%) 14,812 (24.3%) 4,739 (7.8%) 4,739 (7.8%) 1,058 (1.7%) 21,551 (35.4%) 24,395 (40.1%) 19,342 (31.8%) 302 (0.5%) | -0.00 (-0.01, 0.01) -(-, -) -( |
| Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of SPP-4i; n (%) Concomitant use or initiation of SPP-4i; n (%) Concomitant use or initiation of SPP-4i; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Insulins; n (%) Past use of Insulins; n (%) Past use of Sulfonylureas; n (%) Past use of Sulfonylureas; n (%) Past use of SPP-4i; n (% | 212 (0.96) 210 [1.00, 3.00] 1.00, 7.00 61,339 (49.3%) 22,397 (18.0%) 20,237 (16.3%) 24.62 (2.0%) 21,296 (17.1%) 7,079 (5.7%) 81.498 (65.5%) 29,354 (23.6%) 28,787 (23.1%) 4,186 (3.4%) 29,247 (23.5%) 9,773 (7.9%) 90,662 (72.8%) 24.04 (1.9%) 43.619 (35.0%) 53,555 (43.0%) 41,983 (33.7%) 698 (0.6%) 23,870 (19.2%) | 2.08 (0.96) 2.00 [1.00, 3.00] 1.00, 7.00 29,479 (48.3%) 10.552 (17.3%) 8.707 (14.3%) 1.273 (21%) 10.715 (17.5%) 3.381 (5.5%) 39,433 (64.5%) 13,941 (22.8%) 12.606 (20.6%) 2.226 (3.6%) 43,860 (71.8%) 4,756 (7.8%) 43,860 (71.8%) 1,058 (1.7%) 21,633 (35.4%) 24,449 (40.0%) 19,388 (31.7%) 303 (0.5%) 10,613 (17.4%) | 0.04 (0.03, 0.05) -(-,-) -(-,-) 1.0% (0.5%, 1.5%) 0.7% (0.4%, 1.1%) 2.0% (1.7%, 2.4%) -0.1% (-0.2%, 0.0%) -0.4% (-0.8%, -0.1%) 0.2% (-0.1%, 0.4%) 0.2% (-0.5%, 1.4%) 0.8% (0.4%, 1.2%) 2.5% (2.1%, 2.9%) -0.3% (-0.5%, -0.1%) -0.3% (-0.5%, -0.1%) 0.0% (0.5%, 1.4%) 0.8% (0.4%, 1.2%) 2.5% (2.1%, 2.9%) -0.3% (-0.5%, 0.1%) -0.3% (-0.5%, 0.1%) 3.0% (2.5%, 3.5%) 0.4% (-0.8%, 0.1%) 3.0% (2.5%, 3.5%) 2.0% (1.5%, 2.4%) 0.1% (-0.9%, 0.1%) 3.0% (2.5%, 3.5%) | 2.08 (0.95) 2.00 [1.00, 3.00] 1.00, 7.00 29,467 (48.4%) 10.364 (17.0%) 8.702 (14.3%) 1.261 (2.1%) 10,540 (17.3%) 3.342 (5.5%) 3.342 (5.5%) 3.342 (5.5%) 12,605 (20.7%) 12,605 (20.7%) 12,605 (20.7%) 14,735 (24.2%) 4,746 (7.8%) 43,638 (71.7%) 10,68 (1.8%) 21,701 (35.7%) 24,381 (40.1%) 19,378 (31.8%) 19,378 (31.8%) 10,709 (17.6%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,388 (48.3%)<br>10,510 (17.3%)<br>8.694 (14.3%)<br>1,265 (21%)<br>10,665 (17.5%)<br>3,369 (5.5%)<br>33,391 (64.6%)<br>13,881 (22.8%)<br>12,581 (20.7%)<br>2,209 (3.6%)<br>14,812 (24.3%)<br>4,739 (7.8%)<br>4,739 (7.8%)<br>21,551 (35.4%)<br>24,395 (40.1%)<br>19,342 (31.8%)<br>302 (0.5%)<br>10,598 (17.4%) | -0.00 (-0.01, 0.01) -(-, -) -( |
| Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of SPP-4; n (%) Concomitant use or initiation of SPP-4; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformin; n (%) Past use of Metformin; n (%) Past use of SpP-4; n (%) Past use of SpP-4; n (%) Past use of SpP-4; n (%) Past use of SpP-4; n (%) Past use of SpP-4; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE.is/ARB's; n (%) ARN; n (%) Thiazides; n (%) Beta-blockers; n (%) Calcium channel blockers; n (%) Digoxin / Digitoxin; n (%) Other diuretics; n (%) | 212 (0.96) 200 [1.00, 3.00] 1.00, 7.00 61,339 (49.3%) 22,397 (18.0%) 20,237 (16.3%) 24,62 (2.0%) 21,296 (17.1%) 7,079 (5.7%) 31,498 (65.5%) 29,354 (23.6%) 28,787 (23.1%) 4,186 (3.4%) 29,247 (23.5%) 9,773 (7.9%) 90,662 (72.8%) 2,404 (1.9%) 43,619 (35.0%) 53,555 (43.0%) 41,983 (33.7%) 698 (0.6%) 23,870 (19.2%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,479 (48.3%)<br>10,552 (17.3%)<br>8,707 (14.3%)<br>1,273 (21%)<br>10,715 (17.5%)<br>3,381 (5.5%)<br>39,433 (64.5%)<br>13,941 (22.8%)<br>12,606 (20.6%)<br>2,226 (3.6%)<br>4,756 (7.8%)<br>43,860 (71.8%)<br>1,058 (1.7%)<br>21,633 (35.4%)<br>24,449 (40.0%)<br>19,388 (31.7%)<br>303 (0.5%)<br>10,613 (17.4%)<br>5,595 (9.2%) | 0.04 (0.03, 0.05) -(-,-) -(-,-) 1.0% (0.5%, 1.5%) 0.7% (0.4%, 1.1%) 2.0% (1.7%, 2.4%) -0.1% (-0.2%, 0.0%) -0.4% (-0.8%, -0.1%) 0.2% (-0.1%, 0.4%) 0.9% (0.5%, 1.4%) 0.8% (0.5%, 1.4%) 0.8% (0.5%, 1.4%) 0.8% (0.5%, 0.1%) -0.3% (-0.5%, 0.1%) -0.3% (-0.5%, 0.1%) -0.3% (-0.5%, 0.1%) 0.9% (1.3%, -0.5%) 0.1% (-0.2%, 0.3%) 1.0% (0.6%, 1.5%) 0.2% (0.1%, 0.3%) 3.0% (2.5%, 3.5%) 2.0% (1.5%, 2.4%) 0.1% (-0.0%, 0.1%) 1.8% (1.4%, 2.2%) 0.5% (0.2%, 0.8%) | 2.08 (0.95) 2.00 [1.00, 3.00] 1.00, 7.00 29,467 (48.4%) 10,364 (17.0%) 8,702 (14.3%) 1,261 (2.1%) 10,540 (17.3%) 3,342 (5.5%) 33,471 (64.9%) 13,722 (22.6%) 12,605 (20.7%) 2,230 (3.7%) 14,735 (24.2%) 4,746 (7.8%) 43,638 (71.7%) 1,068 (1.8%) 2,1701 (35.7%) 24,381 (40.1%) 19,378 (31.8%) 300 (0.5%) 10,099 (17.6%) 5,639 (9.3%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,388 (48.3%)<br>10,510 (17.3%)<br>8.694 (14.3%)<br>1,265 (21%)<br>10,665 (17.5%)<br>3,369 (5.5%)<br>3,369 (5.5%)<br>13,881 (22.8%)<br>12,581 (20.7%)<br>2,209 (3.6%)<br>14,812 (24.3%)<br>4,739 (7.8%)<br>43,704 (71.8%)<br>10,588 (1.7%)<br>24,395 (40.1%)<br>19,342 (31.8%)<br>302 (0.5%)<br>10,589 (17.4%)<br>5,579 (9.2%) | -0.00 (-0.01, 0.01) -(-, -) -(-, -) -(-, -) -0.2% (-0.7%, 0.2%) -0.2% (-0.7%, 0.2%) -0.0% (-0.4%, 0.4%) -0.0% (-0.2%, 0.2%) -0.2% (-0.6%, 0.2%) -0.3% (-0.3%, 0.2%) -0.3% (-0.3%, 0.2%) -0.3% (-0.3%, 0.2%) -0.0% (-0.4%, 0.5%) -0.0% (-0.4%, 0.5%) -0.0% (-0.4%, 0.5%) -0.0% (-0.6%, 0.4%) -0.1% (-0.6%, 0.4%) -0.1% (-0.6%, 0.4%) -0.0% (-0.3%, 0.3%) -0.1% (-0.6%, 0.5%) -0.0% (-0.5%, 0.6%) -0.0% (-0.5%, 0.6%) -0.0% (-0.5%, 0.6%) -0.0% (-0.5%, 0.6%) -0.0% (-0.1%, 0.1%) |
| Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformir; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of SP-4; n (%) Concomitant use or initiation of PP-4; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformir, n (%) Past use of Metformir, n (%) Past use of SpL1-2; n (%) Past use of SPP-4; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ACE-is/ARB's; n (%) Thiazides; n (%) Calcium channel blockers; n (%) Digoxin / Digitoxin; n (%) Loop diuretics; n (%) Intravenous diuretics; n (%) | 212 (0.96) 200 [1.00, 3.00] 1.00, 7.00 61.339 (49.3%) 22.397 (18.0%) 20.237 (16.3%) 2.462 (2.0%) 21.296 (17.1%) 7.079 (5.7%) 81.498 (65.5%) 29.354 (23.6%) 28.787 (23.1%) 4.186 (3.4%) 29.247 (23.5%) 9.773 (7.9%) 90.662 (72.8%) 2.404 (1.9%) 43.619 (35.0%) 53.555 (43.0%) 41.983 (33.7%) 698 (0.6%) 23.870 (19.2%) 12.049 (9.7%) 1.808 (1.5%) | 2.08 (0.96)<br>2.00 [1.00, 3.00]<br>1.00, 7.00<br>29,479 (48.3%)<br>10.552 (17.3%)<br>8,707 (14.3%)<br>1.273 (21%)<br>10,715 (17.5%)<br>3,381 (5.5%)<br>39,433 (64.5%)<br>12,606 (20.6%)<br>2,226 (3.6%)<br>14,886 (24.4%)<br>4,756 (7.8%)<br>43,860 (71.8%)<br>1,058 (1.7%)<br>21,633 (35.4%)<br>24,449 (40.0%)<br>19,388 (31.7%)<br>303 (0.5%)<br>10,613 (17.4%)<br>5,595 (9.2%)<br>762 (1.2%) | 0.04 (0.03, 0.05) -(-,-) -(-,-) 1.0% (0.5%, 1.5%) 0.7% (0.4%, 1.1%) 2.0% (1.7%, 2.4%) -0.1% (-0.2%, 0.0%) -0.4% (-0.8%, -0.1%) 0.2% (-0.1%, 0.4%) 0.9% (0.5%, 1.4%) 0.9% (0.5%, 1.4%) 0.9% (0.5%, 1.4%) -0.3% (-0.5%, 0.1%) -0.3% (-0.5%, 0.1%) -0.9% (1.3%, -0.5%) 0.1% (-0.2%, 0.3%) 1.0% (0.6%, 1.5%) 0.2% (0.1%, 0.3%) -0.4% (-0.8%, 0.1%) 3.0% (2.5%, 3.5%) 2.0% (1.5%, 2.4%) 0.1% (-0.0%, 0.1%) 1.8% (1.4%, 2.2%) 0.5% (0.2%, 0.8%) 0.5% (0.2%, 0.8%) | 2.08 (0.95) 2.08 (0.95) 1.00, 7.00 29,467 (48.4%) 10,364 (17.0%) 8,702 (14.3%) 1,261 (21%) 10,540 (17.3%) 33.42 (5.5%) 39,471 (64.9%) 13,722 (22.6%) 12,605 (20.7%) 2230 (3.7%) 14,735 (24.2%) 47,746 (7.8%) 43,638 (71.7%) 1,068 (1.8%) 21,701 (35.7%) 24,381 (40.1%) 19,378 (31.8%) 300 (0.5%) 10,709 (17.6%) 5,639 (9.3%) 779 (1.3%) | 2.08 (0.96) 2.08 (0.96) 1.00, 7.00 29,388 (48.3%) 10,510 (17.3%) 8.694 (14.3%) 1.0655 (17.5%) 3.369 (5.5%) 39,301 (64.6%) 13,381 (28.9%) 12,581 (20.7%) 2.209 (3.6%) 14,812 (24.3%) 4,739 (7.8%) 43,704 (71.8%) 1.058 (1.7%) 21,551 (35.4%) 24,395 (40.1%) 19,342 (31.8%) 302 (0.5%) 10,598 (17.4%) 5,579 (9.2%) 759 (1.2%) | -0.00 (-0.01, 0.01) -(-, -) -( |
| Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Sulforulymas; n (%) Concomitant use or initiation of Sulforulymas; n (%) Concomitant use or initiation of Sulforulymas; n (%) Concomitant use or initiation of Sulforulymas; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Insulins; n (%) Past use of Insulins; n (%) Past use of Sulforulymeas; n (%) Past use of Sulforulymeas; n (%) Past use of Sulforulymeas; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARBs; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARBs; n (%) Bata-blockers; n (%) Diazides; n (%) Beta-blockers; n (%) Diazides; n (%) Digoxin / Digitoxin; n (%) Loop diuretics; n (%) Nitrates; n (%) Nitrates; n (%) | 212 (0.96) 210 (1.00, 3.00) 1.00, 7.00 61,339 (49.3%) 22,397 (18.0%) 22,397 (18.0%) 22,397 (18.0%) 24,62 (2.0%) 21,296 (17.1%) 7,079 (5.7%) 81,498 (65.5%) 29,354 (23.6%) 28,787 (23.1%) 41,186 (3.4%) 29,247 (23.5%) 9,773 (7.9%) 90,662 (7.28%) 24,04 (1.28%) 24,04 (1.38%) 43,619 (35.0%) 53,555 (43.0%) 41,983 (33.7%) 698 (0.6%) 23,870 (19.2%) 12,049 (9.7%) 18,088 (1.5%) 8,119 (6.5%) | 2.08 (0.96) 2.00 [1.00, 3.00] 1.00, 7.00 29,479 (48.3%) 10.552 (17.3%) 8.707 (14.3%) 1.273 (21%) 10.715 (17.5%) 3,381 (5.5%) 39,433 (64.5%) 13,941 (22.8%) 12,606 (20.6%) 2.226 (3.6%) 14,886 (24.4%) 4.756 (7.8%) 43,860 (71.8%) 10,58 (1.7%) 21,633 (35.4%) 24,449 (40.0%) 19,388 (31.7%) 303 (0.5%) 10,613 (17.4%) 5,595 (9.2%) 762 (1.2%) 3,410 (5.6%) | 0.04 (0.03, 0.05) -(-,-) -(-,-) -(-,-) 1.0% (0.5%, 1.5%) 0.7% (0.4%, 1.1%) -0.1% (0.4%, 1.1%) -0.1% (-0.2%, 0.0%) -0.4% (-0.8%, -0.1%) 0.2% (-0.1%, 0.4%) 0.8% (0.4%, 1.2%) 2.5% (2.1%, 2.9%) -0.3% (-0.5%, -0.1%) -0.9% (0.5%, -0.1%) -0.9% (1.3%, -0.5%) 1.0% (0.6%, -0.1%) -0.9% (1.3%, -0.5%) -0.4% (-0.8%, 0.1%) -0.9% (1.3%, -0.5%) -0.4% (-0.8%, 0.1%) 3.0% (2.5%, 3.5%) 2.0% (1.5%, 2.4%) 0.1% (-0.9%, 0.1%) 1.8% (1.4%, 2.2%) 0.5% (0.2%, 0.3%) 0.9% (0.7%, 0.3%) | 2.08 (0.95) 2.00 [1.00, 3.00] 1.00, 7.00 29,467 (48.4%) 10.364 (17.0%) 8.702 (14.3%) 1.261 (2.1%) 10.540 (17.3%) 3.342 (5.5%) 39,471 (64.9%) 13,722 (22.6%) 12,605 (20.7%) 2.230 (3.7%) 14,735 (24.2%) 4,746 (7.8%) 43,638 (71.7%) 10,68 (18.%) 21,701 (35.7%) 24,381 (40.1%) 19,378 (31.8%) 300 (0.5%) 10,709 (17.6%) 5,639 (9.3%) 779 (1.3%) 3,384 (5.6%) | 2.08 (0.96) 2.08 (0.96) 2.00 (1.00, 3.00) 1.00, 7.00 29,388 (48.3%) 10.510 (17.3%) 8.694 (14.3%) 1.265 (2.1%) 10.665 (17.5%) 33,665 (5.5%) 33,9301 (64.6%) 13,881 (22.8%) 12,581 (20.7%) 2.209 (3.6%) 14,812 (24.3%) 4,739 (7.8%) 4,739 (7.8%) 10,588 (17.9%) 21,551 (35.4%) 24,395 (40.1%) 19,342 (31.8%) 302 (0.5%) 10,598 (17.4%) 5,579 (9.2%) 759 (1.2%) 3,409 (5.6%) | -0.00 (-0.01, 0.01) -(-, -) -(-, -) -(-, -) -(-, -) -(-, -) -(-, -) -0.2% (-0.7%, 0.2%) -0.2% (-0.7%, 0.2%) -0.2% (-0.6%, 0.2%) -0.2% (-0.6%, 0.2%) -0.0% (-0.2%, 0.2%) -0.0% (-0.3%, 0.2%) -0.3% (-0.3%, 0.2%) -0.3% (-0.3%, 0.2%) -0.3% (-0.3%, 0.3%) -0.3% (-0.3%, 0.3%) -0.1% (-0.6%, 0.4%) -0.0% (-0.3%, 0.3%) -0.1% (-0.6%, 0.4%) -0.0% (-0.6%, 0.5%) -0.0% (-0.6%, 0.5%) -0.0% (-0.6%, 0.5%) -0.0% (-0.5%, 0.6%) -0.0% (-0.1%, 0.1%) -0.2% (-0.2%, 0.6%) -0.9% (-0.1%, 0.1%) |
| Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylures; n (%) Concomitant use or initiation of Sulfonylures; n (%) Concomitant use or initiation of SPP-4i; n (%) Concomitant use or initiation of SPP-4i; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Insulins; n (%) Past use of Insulins; n (%) Past use of Sulfonylureas; n (%) Past use of Sulfonylureas; n (%) Past use of SPP-4i; | 212 (0.96) 210 (1.00, 3.00) 1.00, 7.00 61,339 (49.3%) 22,397 (18.0%) 20,237 (16.3%) 24.62 (2.0%) 21,296 (17.1%) 7,079 (5.7%) 81.498 (65.5%) 29,354 (23.6%) 28,787 (23.1%) 4,186 (3.4%) 29,247 (23.5%) 9,773 (7.9%) 90,662 (72.8%) 24.04 (1.9%) 43.619 (35.0%) 53,555 (43.0%) 41,983 (33.7%) 698 (0.6%) 23,870 (19.2%) 12,049 (9.7%) 1.808 (1.5%) 8,119 (6.5%) 1,076 (2.5%) | 2.08 (0.96) 2.00 [1.00, 3.00] 1.00, 7.00 29,479 (48.3%) 10,552 (17.3%) 8.707 (14.3%) 1,273 (21%) 10,715 (17.5%) 3,381 (5.5%) 39,433 (64.5%) 13,941 (22.8%) 12,606 (20.6%) 2,226 (3.6%) 43,860 (71.8%) 4,756 (7.8%) 43,860 (71.8%) 1,058 (1.7%) 21,633 (35.4%) 24,449 (40.0%) 19,388 (31.7%) 303 (0.5%) 10,613 (17.4%) 5,595 (9.2%) 762 (1.2%) 3,410 (5.6%) 1,374 (2.2%) | 0.04 (0.03, 0.05) -(-,-) -(-,-) 1.0% (0.5%, 1.5%) 0.7% (0.4%, 1.1%) 2.0% (1.7%, 2.4%) -0.1% (-0.2%, 0.0%) -0.4% (-0.8%, -0.1%) 0.2% (-0.1%, 0.4%) 0.8% (0.4%, 1.2%) 2.5% (2.1%, 2.9%) -0.3% (-0.5%, -0.1%) -0.3% (-0.5%, -0.1%) 0.9% (0.5%, 1.4%) 0.8% (0.4%, 1.2%) 2.5% (2.1%, 2.9%) -0.3% (-0.5%, 0.1%) -0.3% (-0.5%, 0.1%) -0.9% (-1.3%, -0.5%) 0.1% (-0.2%, 0.3%) 1.0% (0.5%, 1.5%) 0.2% (0.1%, 0.3%) -0.4% (-0.9%, 0.1%) 3.0% (2.5%, 3.5%) 2.0% (1.5%, 2.4%) 0.1% (-0.0%, 0.1%) 1.9% (-0.0%, 0.1%) 0.5% (0.2%, 0.8%) 0.2% (0.1%, 0.3%) 0.9% (0.7%, 1.2%) | 2.08 (0.95) 2.08 (0.95) 1.00, 7.00 2.9,467 (48.4%) 10.364 (17.0%) 8.702 (14.3%) 1.261 (2.1%) 10,540 (17.3%) 3.342 (5.5%) 3.342 (5.5%) 12,605 (20.7%) 12,701 (35.7%) 14,735 (24.2%) 4,746 (7.8%) 43,638 (71.7%) 10,68 (1.8%) 21,701 (35.7%) 24,381 (40.1%) 19,378 (31.8%) 300 (0.5%) 10,709 (17.6%) 5,639 (9.3%) 779 (1.3%) 3,384 (5.6%) 1,337 (2.2%) | 2.08 (0.96) 2.08 (0.96) 1.00, 7.00 29,388 (48.3%) 10,510 (17.3%) 8.694 (14.3%) 1,265 (21%) 10,665 (17.5%) 3,369 (5.5%) 33,393 (164.6%) 13,881 (22.8%) 12,581 (20.7%) 2,209 (3.6%) 14,812 (24.3%) 4,739 (7.8%) 4,739 (7.8%) 24,395 (40.1%) 19,342 (31.8%) 302 (0.5%) 10,598 (17.4%) 5,579 (1.2%) 3,409 (5.6%) 1,371 (2.3%) | -0.00 (-0.01, 0.01) -(-, -) -( |
| Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformir; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of SP-4; n (%) Concomitant use or initiation of SP-4; n (%) Concomitant use or initiation of SP-4; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformir, n (%) Past use of Metformir, n (%) Past use of Sulfonylureas; n (%) Past use of SPP-4; n (%) Past use of Sulfonylureas; n (%) Past use of SPP-4; n (%) Past use | 212 (0.96) 200 [1.00, 3.00] 1.00, 7.00 61.339 (49.3%) 22.397 (18.0%) 20.237 (16.3%) 24.62 (2.0%) 21.296 (17.1%) 7.079 (5.7%) 81.498 (65.5%) 29.354 (23.6%) 28.787 (23.1%) 4.186 (3.4%) 29.247 (23.5%) 9.773 (7.9%) 90.662 (72.8%) 2404 (1.9%) 43.619 (35.0%) 53.555 (43.0%) 41.983 (33.7%) 698 (0.5%) 23.870 (19.2%) 12.049 (9.7%) 1.808 (1.5%) 8.119 (6.5%) 99.996 (80.3%) 17.009 (13.7%) | 2.08 (0.96) 2.00 [1.00, 3.00] 1.00, 7.00 29,479 (48.3%) 10.552 (17.3%) 8,707 (14.3%) 10.715 (17.5%) 3,381 (5.5%) 39,433 (64.5%) 12,606 (20.6%) 2,226 (3.6%) 14,886 (24.4%) 4,756 (7.8%) 43,860 (71.8%) 1,058 (1.7%) 21,633 (35.4%) 24,449 (40.0%) 19,388 (31.7%) 303 (0.5%) 10,613 (17.4%) 5,595 (9.2%) 762 (1.2%) 3,410 (5.6%) 1,374 (2.2%) 47,091 (77.1%) 8,538 (14.0%) | 0.04 (0.03, 0.05) -(-,-) -(-,-) 1.0% (0.5%, 1.5%) 0.7% (0.4%, 1.1%) 2.0% (1.7%, 2.4%) -0.1% (-0.2%, 0.0%) -0.4% (-0.8%, -0.1%) 0.2% (-0.1%, 0.4%) 0.9% (0.5%, 1.4%) 0.9% (0.5%, 1.4%) 0.9% (0.5%, 1.4%) -0.3% (-0.5%, -0.1%) -0.3% (-0.5%, -0.1%) -0.9% (1.3%, -0.5%) 0.1% (-0.2%, 0.3%) 1.0% (0.6%, 1.5%) 0.2% (0.1%, 0.3%) -0.4% (-0.8%, 0.1%) 3.0% (2.5%, 3.5%) 2.0% (1.5%, 2.4%) 0.1% (-0.0%, 0.1%) 1.8% (1.4%, 2.2%) 0.2% (0.1%, 0.3%) 0.2% (0.1%, 0.3%) 0.2% (0.1%, 0.3%) 0.2% (0.1%, 0.3%) | 2.08 (0.95) 2.08 (0.95) 1.00, 7.00 2.9.467 (48.4%) 10.364 (17.0%) 8.702 (14.3%) 1.0540 (17.3%) 3.342 (5.5%) 39.471 (64.9%) 13,722 (22.6%) 12,605 (20.7%) 2.230 (3.7%) 14,735 (24.2%) 4,746 (7.8%) 43,638 (71.7%) 1.068 (1.8%) 21,701 (35.7%) 24,381 (40.1%) 19,378 (31.8%) 300 (0.5%) 10,099 (17.6%) 5,639 (9.3%) 779 (1.3%) 3.384 (5.6%) 1.384 (5.6%) 1.387 (22.9%) 4.6,959 (77.2%) 8,550 (14.1%) | 2.08 (0.96) 2.08 (0.96) 2.00 [1.00, 3.00] 1.00, 7.00 29,388 (48.3%) 10,510 (17.3%) 8.694 (14.3%) 1.265 (21%) 10,665 (17.5%) 33,301 (64.6%) 13,381 (28.8%) 12,581 (20.7%) 2.209 (3.6%) 14,812 (24.3%) 4,739 (7.8%) 43,704 (71.8%) 1.058 (1.7%) 21,551 (35.4%) 24,395 (40.1%) 19,342 (31.8%) 302 (0.5%) 10,598 (17.4%) 5,579 (9.2%) 759 (1.2%) 3,409 (5.6%) 1,371 (2.3%) 46,986 (77.2%) 8,507 (14.0%) | -0.00 (-0.01, 0.01) -(-, -) -( |
| Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of SGLT-2i; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Insulins; n (%) Past use of Insulins; n (%) Past use of Insulins; n (%) Past use of SQLT-2i; n (%) Past use of SQLT-2i; n (%) Past use of Any other glucose-lowering drugs; n (%) Past use of Any other glucose-lowering drugs; n (%) Past use of Any other glucose-lowering drugs; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARBs; n (%) ARNI; n (%) Thiazides; n (%) Beta-blockers; n (%) Digoxin / Digitoxin; n (%) Digoxin / Digitoxin; n (%) Loop diuretics; n (%) Intravenous diuretics; n (%) Nitrates; n (%) Anti-arrhythmics; n (%) Statins; n (%) Anti-arrhythmics and other lipid-lowering drugs; n (%) Anti-arrhythmics and other lipid-lowering drugs; n (%) Anti-arrhythmics and other lipid-lowering drugs; n (%) | 212 (0.96) 210 (1.00, 3.00) 1.00, 7.00 61,339 (49.3%) 22,397 (18.0%) 22,397 (18.0%) 22,397 (18.0%) 24,62 (2.0%) 21,296 (17.1%) 7,079 (5.7%) 81,498 (65.5%) 29,354 (23.6%) 28,787 (23.1%) 41,186 (3.4%) 29,247 (23.5%) 9,773 (7.9%) 90,662 (72.8%) 24,04 (1.9%) 43,619 (35.0%) 53,555 (43.0%) 41,983 (33.7%) 698 (0.6%) 23,870 (19.2%) 12,049 (9.7%) 12,049 (9.7%) 18.19 (6.5%) 3,076 (2.5%) 99,996 (80.3%) 17,009 (13.7%) 12,657 (10.2%) | 2.08 (0.96) 2.00 [1.00, 3.00] 1.00, 7.00 29,479 (48.3%) 10.552 (17.3%) 8.707 (14.3%) 1.273 (21%) 10.715 (17.5%) 3,381 (5.5%) 39,433 (64.5%) 13,941 (22.8%) 12,606 (20.6%) 2.226 (3.6%) 14,886 (24.4%) 4.756 (7.8%) 43,860 (71.8%) 10,58 (1.7%) 21,633 (35.4%) 24,449 (40.0%) 19,388 (31.7%) 303 (0.5%) 10,613 (17.4%) 5,595 (9.2%) 762 (1.2%) 3,410 (5.6%) 1,374 (2.2%) 47,091 (77.1%) 8,538 (14.0%) 5,400 (8.8%) | 0.04 (0.03, 0.05) -(-,-) -(-,-) -(-,-) -(-,-) 1.0% (0.5%, 1.5%) 0.7% (0.4%, 1.1%) 2.0% (1.7%, 2.4%) -0.1% (-0.2%, 0.0%) -0.4% (-0.8%, -0.1%) 0.2% (-0.1%, 0.4%) 0.8% (0.4%, 1.2%) 2.5% (2.1%, 2.9%) -0.3% (-0.5%, -0.1%) 0.9% (0.5%, 1.4%) 0.8% (0.4%, 1.2%) 2.5% (2.1%, 2.9%) -0.3% (-0.5%, -0.1%) -0.9% (1.3%, -0.5%) 1.0% (0.6%, -0.1%) 3.0% (2.5%, 3.5%) 2.0% (1.5%, 2.4%) 0.1% (-0.0%, 0.1%) 1.8% (1.4%, 2.2%) 0.5% (0.2%, 0.3%) 0.9% (0.7%, 1.2%) 0.9% (0.1%, 0.3%) 0.9% (0.7%, 1.2%) 0.9% (0.1%, 0.3%) 0.9% (0.7%, 1.2%) 0.2% (0.1%, 0.3%) 0.9% (0.7%, 1.2%) 0.2% (0.1%, 0.3%) | 2.08 (0.95) 2.08 (0.95) 1.00, 7.00 2.9.467 (48.4%) 10.364 (17.0%) 8.702 (14.3%) 1.261 (2.1%) 10.540 (17.3%) 3.342 (5.5%) 39.471 (64.9%) 13.722 (22.6%) 12.605 (20.7%) 2.230 (3.7%) 14.735 (24.2%) 4.746 (7.8%) 4.746 (7.8%) 4.3638 (71.7%) 1.068 (18%) 21.701 (35.7%) 24.381 (40.1%) 19.378 (31.8%) 300 (0.5%) 10.709 (17.6%) 5.639 (9.3%) 779 (1.3%) 3.384 (5.6%) 1.337 (2.2%) 4.6.959 (77.2%) 8.550 (14.1%) 5.5427 (8.9%) | 2.08 (0.96) 2.08 (0.96) 2.00 [1.00, 3.00] 1.00, 7.00 29,388 (48.3%) 10.510 (17.3%) 8.694 (14.3%) 1.265 (2.1%) 10.665 (17.5%) 33,695 (5.5%) 39,301 (64.6%) 13,881 (22.8%) 12,581 (20.7%) 2.209 (3.6%) 14,812 (24.3%) 4,739 (7.8%) 4,739 (7.8%) 4,739 (7.8%) 21,551 (35.4%) 24,395 (40.1%) 19,342 (31.8%) 302 (0.5%) 10,598 (17.4%) 5,579 (9.2%) 759 (12.9%) 3,409 (5.6%) 1,371 (2.3%) 46,986 (77.2%) 8,507 (14.0%) 5,395 (8.9%) | -0.00 (-0.01, 0.01) -(-, -) -( |
| Number of antidiabetic drugs on CEDmean (sd)median [IQR]min, max Concomitant use or initiation of Metformir; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of SP-4; n (%) Concomitant use or initiation of SP-4; n (%) Concomitant use or initiation of SP-4; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformir, n (%) Past use of Metformir, n (%) Past use of Sulfonylureas; n (%) Past use of SPP-4; n (%) Past use of Sulfonylureas; n (%) Past use of SPP-4; n (%) Past use | 212 (0.96) 200 [1.00, 3.00] 1.00, 7.00 61.339 (49.3%) 22.397 (18.0%) 20.237 (16.3%) 24.62 (2.0%) 21.296 (17.1%) 7.079 (5.7%) 81.498 (65.5%) 29.354 (23.6%) 28.787 (23.1%) 4.186 (3.4%) 29.247 (23.5%) 9.773 (7.9%) 90.662 (72.8%) 2404 (1.9%) 43.619 (35.0%) 53.555 (43.0%) 41.983 (33.7%) 698 (0.5%) 23.870 (19.2%) 12.049 (9.7%) 1.808 (1.5%) 8.119 (6.5%) 99.996 (80.3%) 17.009 (13.7%) | 2.08 (0.96) 2.00 [1.00, 3.00] 1.00, 7.00 29,479 (48.3%) 10.552 (17.3%) 8,707 (14.3%) 10.715 (17.5%) 3,381 (5.5%) 39,433 (64.5%) 12,606 (20.6%) 2,226 (3.6%) 14,886 (24.4%) 4,756 (7.8%) 43,860 (71.8%) 1,058 (1.7%) 21,633 (35.4%) 24,449 (40.0%) 19,388 (31.7%) 303 (0.5%) 10,613 (17.4%) 5,595 (9.2%) 762 (1.2%) 3,410 (5.6%) 1,374 (2.2%) 47,091 (77.1%) 8,538 (14.0%) | 0.04 (0.03, 0.05) -(-,-) -(-,-) 1.0% (0.5%, 1.5%) 0.7% (0.4%, 1.1%) 2.0% (1.7%, 2.4%) -0.1% (-0.2%, 0.0%) -0.4% (-0.8%, -0.1%) 0.2% (-0.1%, 0.4%) 0.9% (0.5%, 1.4%) 0.9% (0.5%, 1.4%) 0.9% (0.5%, 1.4%) -0.3% (-0.5%, -0.1%) -0.3% (-0.5%, -0.1%) -0.9% (1.3%, -0.5%) 0.1% (-0.2%, 0.3%) 1.0% (0.6%, 1.5%) 0.2% (0.1%, 0.3%) -0.4% (-0.8%, 0.1%) 3.0% (2.5%, 3.5%) 2.0% (1.5%, 2.4%) 0.1% (-0.0%, 0.1%) 1.8% (1.4%, 2.2%) 0.2% (0.1%, 0.3%) 0.2% (0.1%, 0.3%) 0.2% (0.1%, 0.3%) 0.2% (0.1%, 0.3%) | 2.08 (0.95) 2.08 (0.95) 1.00, 7.00 2.9.467 (48.4%) 10.364 (17.0%) 8.702 (14.3%) 1.0540 (17.3%) 3.342 (5.5%) 39.471 (64.9%) 13,722 (22.6%) 12,605 (20.7%) 2.230 (3.7%) 14,735 (24.2%) 4,746 (7.8%) 43,638 (71.7%) 1.068 (1.8%) 21,701 (35.7%) 24,381 (40.1%) 19,378 (31.8%) 300 (0.5%) 10,099 (17.6%) 5,639 (9.3%) 779 (1.3%) 3.384 (5.6%) 1.384 (5.6%) 1.387 (22.9%) 4.6,959 (77.2%) 8,550 (14.1%) | 2.08 (0.96) 2.08 (0.96) 2.00 [1.00, 3.00] 1.00, 7.00 29,388 (48.3%) 10,510 (17.3%) 8.694 (14.3%) 1.265 (21%) 10,665 (17.5%) 33,301 (64.6%) 13,381 (28.8%) 12,581 (20.7%) 2.209 (3.6%) 14,812 (24.3%) 4,739 (7.8%) 43,704 (71.8%) 1.058 (1.7%) 21,551 (35.4%) 24,395 (40.1%) 19,342 (31.8%) 302 (0.5%) 10,598 (17.4%) 5,579 (9.2%) 759 (1.2%) 3,409 (5.6%) 1,371 (2.3%) 46,986 (77.2%) 8,507 (14.0%) | -0.00 (-0.01, 0.01) -(-, -) -( |

| i | | | | _ | | |
|---|---|---|---|---|---|---|
| NSAIDS; n (%) | 42,649 (34.3%) | 20,682 (33.9%) | 0.4% (-0.0%, 0.9%) | 20,658 (34.0%) | 20,620 (33.9%) | 0.1% (-0.5%, 0.6%) |
| Oral corticosteroids; n (%) | 32,991 (26.5%) | 17,020 (27.9%) | -1.4% (-1.8%, -0.9%) | 17,052 (28.0%) | 16,929 (27.8%) | 0.2% (-0.3%, 0.7%) |
| Osteoporosis agents (incl. bisphosphonates); n (%) | 3,548 (2.9%) | 1,450 (2.4%) | 0.5% (0.3%, 0.6%) | 1,460 (2.4%) | 1,450 (2.4%) | 0.0% (-0.2%, 0.2%) |
| Opioids; n (%) | 39,602 (31.8%) | 18,894 (30.9%) | 0.9% (0.4%, 1.3%) | 18,757 (30.8%) | 18,844 (31.0%) | -0.1% (-0.7%, 0.4%) |
| Anti-depressants; n (%) | 50,810 (40.8%) | 24,541 (40.2%) | 0.7% (0.2%, 1.1%) | 24,510 (40.3%) | 24,456 (40.2%) | 0.1% (-0.5%, 0.6%) |
| Antipsychotics; n (%) | 6,244 (5.0%) | 2,823 (4.6%) | 0.4% (0.2%, 0.6%) | 2,827 (4.6%) | 2,812 (4.6%) | 0.0% (-0.2%, 0.3%) |
| Anxiolytics / hypnotics, benzos; n (%) | 27,986 (22.5%) | 13,879 (22.7%) | -0.2% (-0.6%, 0.2%) | 13,808 (22.7%) | 13,822 (22.7%) | -0.0% (-0.5%, 0.4%) |
| Dementia medications; n (%) | 1,722 (1.4%) | 640 (1.0%) | 0.3% (0.2%, 0.4%) | 609 (1.0%) | 640 (1.1%) | -0.1% (-0.2%, 0.1%) |
| Urinary tract infections antibiotics; n (%) | 58,613 (47.1%) | 29,223 (47.8%) | -0.7% (-1.2%, -0.3%) | 28,977 (47.6%) | 29,096 (47.8%) | -0.2% (-0.8%, 0.4%) |
| Laxatives; n (%) | 4,583 (3.7%) | 2,158 (3.5%) | 0.1% (-0.0%, 0.3%) | 2,128 (3.5%) | 2,152 (3.5%) | -0.0% (-0.2%, 0.2%) |
| Number of distinct medications | | | | | | |
| mean (sd) | 14.84 (7.08) | 14.52 (7.22) | 0.32 (0.25, 0.39) | 14.50 (7.13) | 14.53 (7.22) | -0.02 (-0.10, 0.06) |
| median [IOR] | 14.00 [10.00, 19.00] | 13.00 [9.00, 18.00] | - (-, -) | 13.00 [9.00, 18.00] | 13.00 [9.00, 18.00] | - (-, -) |
| min, max | 1.00, 72.00 | 1.00, 69.00 | - (-, -) | 1.00, 72.00 | 1.00, 69.00 | - (-, -) |
| Number of office visits | 100,72.00 | 100,00.00 | ( , , | 100,72100 | 2.00, 05.00 | (, / |
| mean (sd) | 9.85 (7.15) | 9.67 (7.18) | 0.18 (0.11, 0.25) | 9.64 (7.18) | 9.67 (7.17) | -0.03 (-0.11, 0.05) |
| median [IQR] | 8.00 [5.00, 13.00] | 8.00 [5.00, 13.00] | - (-, -) | 8.00 [5.00, 13.00] | 8.00 [5.00, 13.00] | -(-, -) |
| | | | - (-, -)<br>- (-, -) | 0.00, 284.00 | 0.00, 93.00 | 177 |
| min, max | 0.00, 284.00 | 0.00, 93.00 | - (-, -) | 0.00, 284.00 | 0.00, 93.00 | - (-, -) |
| Number of endocrinologist visits | | | | | | |
| mean (sd) | 0.41 (1.36) | 0.43 (1.40) | -0.02 (-0.04, -0.01) | 0.42 (1.41) | 0.43 (1.40) | -0.01 (-0.02, 0.01) |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) |
| min, max | 0.00, 53.00 | 0.00, 85.00 | - (-, -) | 0.00, 53.00 | 0.00, 85.00 | - (-, -) |
| Number of cardiologist visits | 1 | | | ļ | | |
| mean (sd) | 1.64 (3.65) | 1.47 (3.24) | 0.17 (0.13, 0.20) | 1.47 (3.23) | 1.47 (3.25) | -0.00 (-0.04, 0.04) |
| median [IQR] | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | - (-, -) | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | - (-, -) |
| min, max | 0.00, 160.00 | 0.00, 96.00 | - (-, -) | 0.00, 119.00 | 0.00, 96.00 | - (-, -) |
| Number of internal/family medicine visits | | | | | | |
| mean (sd) | 7.32 (8.56) | 6.68 (7.45) | 0.64 (0.56, 0.72) | 6.64 (7.33) | 6.69 (7.46) | -0.05 (-0.13, 0.03) |
| median [IQR] | 5.00 [3.00, 9.00] | 5.00 [3.00, 8.00] | - (-, -) | 5.00 [3.00, 8.00] | 5.00 [3.00, 8.00] | - (-, -) |
| min, max | 0.00, 233.00 | 0.00, 225.00 | - (-, -) | 0.00, 233.00 | 0.00, 225.00 | - (-, -) |
| Number of electrocardiograms (ECG/EKG) | | | | | | |
| mean (sd) | 0.97 (1.68) | 0.89 (1.59) | 0.08 (0.06, 0.10) | 0.89 (1.54) | 0.89 (1.60) | -0.00 (-0.02, 0.02) |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | - (-, -) | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | - (-, -) |
| min, max | 0.00, 52.00 | 0.00, 59.00 | - (-, -) | 0.00, 29.00 | 0.00,59.00 | - (-, -) |
| Number of echocardiograms | 0.00, 32.00 | 0.00, 33.00 | - (-, -) | 0.00, 23.00 | 0.00, 33.00 | - (-, -) |
| mean (sd) | 0.28 (0.64) | 0.25 (0.60) | 0.03 (0.02, 0.04) | 0.25 (0.59) | 0.25 (0.60) | -0.00 (-0.01, 0.01) |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) |
| min, max | 0.00, 15.00 | 0.00, 13.00 | - (-, -) | 0.00, 14.00 | 0.00, 13.00 | - (-, -) |
| Out-of-pocket medication cost | | | | | | |
| mean (sd) | 597.61 (783.11) | 595.25 (793.96) | 2.36 (-5.30, 10.01) | 589.69 (795.01) | 595.59 (794.59) | -5.90 (-14.83, 3.03) |
| median [IQR] | 340.79 [133.09, 792.50] | 340.16 [124.64, 792.59] | - (-, -) | 336.47 [131.17, 778.21] | 340.33 [124.81, 793.12] | - (-, -) |
| min, max | 0.00, 40,518.11 | 0.00, 36,280.29 | - (-, -) | 0.00, 40,518.11 | 0.00, 36,280.29 | - (-, -) |
| Unique brand medicines | | | | | | |
| mean (sd) | 15.12 (7.31) | 14.75 (7.43) | 0.37 (0.30, 0.44) | 14.73 (7.33) | 14.76 (7.43) | -0.02 (-0.11, 0.06) |
| median [IQR] | 14.00 [10.00, 19.00] | 14.00 [9.00, 19.00] | - (-, -) | 14.00 [9.00, 19.00] | 14.00 [9.00, 19.00] | - (-, -) |
| min, max | 1.00, 84.00 | 1.00, 77.00 | - (-, -) | 1.00, 84.00 | 1.00, 77.00 | - (-, -) |
| Unique generic medicines | | | | | | |
| mean (sd) | 14.84 (7.08) | 14.52 (7.22) | 0.32 (0.25, 0.39) | 14.50 (7.13) | 14.53 (7.22) | -0.02 (-0.10, 0.06) |
| median [IOR] | 14.00 [10.00, 19.00] | 13.00 [9.00, 18.00] | - (-, -) | 13.00 [9.00, 18.00] | 13.00 [9.00, 18.00] | - (-, -) |
| min, max | 1.00, 72.00 | 1.00, 69.00 | - (-, -) | 1.00, 72.00 | 1.00, 69.00 | - (-, -) |
| Colonoscopy Sigmoidoscopy; n (%) | 13,600 (10.9%) | 6,647 (10.9%) | 0.0% (-0.3%, 0.3%) | 6,637 (10.9%) | 6,621 (10.9%) | 0.0% (-0.3%, 0.4%) |
| Flu Pneumococcal vaccine; n (%) | 40,282 (32.4%) | 18,348 (30.0%) | 2.3% (1.9%, 2.8%) | 18,317 (30.1%) | 18,307 (30.1%) | 0.0% (-0.5%, 0.5%) |
| Pap smear; n (%) | 8,575 (6.9%) | 4,843 (7.9%) | -1.0% (-1.3%, -0.8%) | 4,779 (7.9%) | 4,791 (7.9%) | -0.0% (-0.3%, 0.3%) |
| PSA test; n(%) | 27,398 (22.0%) | 13,951 (22.8%) | -0.8% (-1.2%, -0.4%) | 13,936 (22.9%) | 13,903 (22.8%) | 0.1% (-0.4%, 0.5%) |
| Fecal occult blood test; n (%) | 5,260 (4.2%) | 2,265 (3.7%) | 0.5% (0.3%, 0.7%) | 2,270 (3.7%) | 2,263 (3.7%) | 0.1% (-0.4%, 0.5%) |
| | 9.938 (8.0%) | 4,505 (3.7%) | 0.5% (0.3%, 0.7%) | 4.519 (7.4%) | 4.501 (7.4%) | 0.0% (-0.2%, 0.2%) |
| Bone mineral density tests; n (%) | | | | | | |
| Mammograms; n (%) | 34,466 (27.7%) | 16,714 (27.4%) | 0.3% (-0.1%, 0.8%) | 16,508 (27.1%) | 16,675 (27.4%) | -0.3% (-0.8%, 0.2%) |
| Telemedicine; n (%) | 29,839 (24.0%) | 14,493 (23.7%) | 0.2% (-0.2%, 0.7%) | 14,378 (23.6%) | 14,412 (23.7%) | -0.1% (-0.5%, 0.4%) |
| HbA1c tests | | | | ļ | | |
| mean (sd) | 2.34 (1.32) | 2.31 (1.32) | 0.03 (0.01, 0.04) | 2.31 (1.35) | 2.31 (1.32) | 0.00 (-0.01, 0.02) |
| | | | - (-, -) | 2.00 [1.00, 3.00] | 2.00 [1.00, 3.00] | - (-, -) |
| median [IQR] | 2.00 [1.00, 3.00] | 2.00 [1.00, 3.00] | | | | |
| median [IQR]min, max | 2.00 [1.00, 3.00]<br>0.00, 75.00 | 2.00 [1.00, 3.00]<br>0.00, 44.00 | - (-, -) | 0.00, 75.00 | 0.00, 44.00 | - (-, -) |
| | | | | | 0.00, 44.00 | - (-, -) |
| min, max | | | | | 0.00, 44.00<br>1.65 (1.14) | 0.00 (-0.01, 0.02) |
| min, max<br>Lipid panels | 0.00, 75.00 | 0.00, 44.00 | - (-, -) | 0.00, 75.00 | | |
| min, max Lipid panelsmean (sd) | 0.00, 75.00<br>1.63 (1.18) | 0.00, 44.00<br>1.65 (1.14) | -(-, -)<br>-0.02 (-0.03, -0.01) | 0.00, 75.00<br>1.65 (1.22) | 1.65 (1.14) | |

| | | | | I | | |
|---|---|---|---|---|---|---|
| Creatinine tests | 2.01 (2.00) | 270 (2.00) | 0.15 (0.10, 0.17) | 2.77 (2.70) | 270 (202) | 0.01 / 0.02 0.04) |
| mean (sd) | 2.91 (2.89) | 2.76 (2.82) | 0.15 (0.12, 0.17) | 2.77 (2.70) | 2.76 (2.82) | 0.01 (-0.03, 0.04) |
| median [IQR] | 2.00 [1.00, 4.00] | 2.00 [1.00, 4.00] | - (-, -) | 2.00 [1.00, 4.00] | 2.00 [1.00, 4.00] | - (-, -) |
| min, max | 0.00, 96.00 | 0.00, 105.00 | - (-, -) | 0.00, 96.00 | 0.00, 105.00 | - (-, -) |
| Natriuretic peptide tests | | | | | | |
| mean (sd) | 0.19 (0.79) | 0.17 (0.68) | 0.02 (0.01, 0.03) | 0.17 (0.69) | 0.17 (0.68) | 0.00 (-0.01, 0.01) |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) |
| min, max | 0.00, 77.00 | 0.00, 28.00 | - (-, -) | 0.00, 55.00 | 0.00, 28.00 | - (-, -) |
| Urine tests | | | | | | |
| mean (sd) | 1.05 (1.64) | 1.03 (1.62) | 0.03 (0.01, 0.04) | 1.03 (1.63) | 1.03 (1.62) | 0.00 (-0.02, 0.02) |
| median [IQR] | 0.00 [0.00, 2.00] | 0.00 [0.00, 1.00] | - (-, -) | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | - (-, -) |
| min, max | 0.00, 66.00 | 0.00, 37.00 | - (-, -) | 0.00, 66.00 | 0.00, 37.00 | - (-, -) |
| Combined comorbidity score | | | | | | |
| mean (sd) | 2.00 (2.40) | 1.79 (2.26) | 0.21 (0.19, 0.24) | 1.78 (2.24) | 1.79 (2.27) | -0.01 (-0.03, 0.02) |
| median [IQR] | 1.00 [0.00, 3.00] | 1.00 [0.00, 3.00] | - (-, -) | 1.00 [0.00, 3.00] | 1.00 [0.00, 3.00] | - (-, -) |
| min, max | -2.00, 17.00 | -2.00, 16.00 | - (-, -) | -2.00, 16.00 | -2.00, 16.00 | - (-, -) |
| Frailty Score | | | | | | |
| mean (sd) | 0.17 (0.06) | 0.16 (0.05) | 0.00 (0.00, 0.00) | 0.16 (0.05) | 0.16 (0.05) | -0.00 (-0.00, 0.00) |
| median [IQR] | 0.16 [0.13, 0.19] | 0.15 [0.13, 0.19] | - (-, -) | 0.15 [0.13, 0.19] | 0.15 [0.13, 0.19] | - (-, -) |
| min, max | 0.03, 0.59 | 0.04, 0.62 | - (-, -) | 0.03, 0.59 | 0.04, 0.62 | - (-, -) |
| Number of Hospitalizations | | | | | | |
| mean (sd) | 0.20 (0.68) | 0.16 (0.57) | 0.04 (0.03, 0.04) | 0.16 (0.57) | 0.16 (0.57) | -0.00 (-0.01, 0.00) |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) |
| min, max | 0.00, 26.00 | 0.00, 12.00 | - (-, -) | 0.00, 22.00 | 0.00, 12.00 | - (-, -) |
| Any hospitalization within prior 91 days; n (%) | 5,303 (4.3%) | 2,136 (3.5%) | 0.8% (0.6%, 0.9%) | 2,079 (3.4%) | 2,131 (3.5%) | -0.1% (-0.3%, 0.1%) |
| Any hospitalization within prior 92-365 days; n (%) | 12,422 (10.0%) | 5,278 (8.6%) | 1.3% (1.1%, 1.6%) | 5,201 (8.5%) | 5,268 (8.7%) | -0.1% (-0.4%, 0.2%) |
| Number of hospitalizations (0, 1, 2 or more) | | | | | | |
| < 1; n (%) | 108,772 (87.4%) | 54,460 (89.1%) | -1.8% (-2.1%, -1.4%) | 54,324 (89.3%) | 54,231 (89.1%) | 0.2% (-0.2%, 0.5%) |
| 1 - <2; n (%) | 10,816 (8.7%) | 4,723 (7.7%) | 1.0% (0.7%, 1.2%) | 4,646 (7.6%) | 4,710 (7.7%) | -0.1% (-0.4%, 0.2%) |
| >= 2; n (%) | 4,882 (3.9%) | 1,909 (3.1%) | 0.8% (0.6%, 1.0%) | 1,878 (3.1%) | 1,907 (3.1%) | -0.0% (-0.2%, 0.1%) |
| Heart failure hospitalization; n (%) | 4,506 (3.6%) | 1,728 (2.8%) | 0.8% (0.6%, 1.0%) | 1,683 (2.8%) | 1,727 (2.8%) | -0.1% (-0.3%, 0.1%) |
| ED visit; n (%) | 36,192 (29.1%) | 16,007 (26.2%) | 2.9% (2.4%, 3.3%) | 15,979 (26.3%) | 15,975 (26.3%) | 0.0% (-0.5%, 0.5%) |
| Acute MI; n (%) | 1,418 (1.1%) | 490 (0.8%) | 0.3% (0.2%, 0.4%) | 505 (0.8%) | 490 (0.8%) | 0.0% (-0.1%, 0.1%) |
| Old MI; n (%) | 5,397 (4.3%) | 2,235 (3.7%) | 0.7% (0.5%, 0.9%) | 2,288 (3.8%) | 2,232 (3.7%) | 0.1% (-0.1%, 0.3%) |
| Heart failure; n (%) | 17,834 (14.3%) | 7,465 (12.2%) | 2.1% (1.8%, 2.4%) | 7,454 (12.3%) | 7,460 (12.3%) | -0.0% (-0.4%, 0.4%) |
| Acute heart failure; n (%) | 4,282 (3.4%) | 1,697 (2.8%) | 0.7% (0.5%, 0.8%) | 1,685 (2.8%) | 1,697 (2.8%) | -0.0% (-0.2%, 0.2%) |
| Microalbuminuria or proteinuria; n (%) | 8,134 (6.5%) | 3,741 (6.1%) | 0.4% (0.2%, 0.6%) | 3,698 (6.1%) | 3,731 (6.1%) | -0.1% (-0.3%, 0.2%) |
| Ratio of brand to generic medications | | | | | | |
| mean (sd) | 1.02 (0.04) | 1.01 (0.04) | 0.00 (0.00, 0.00) | 1.01 (0.04) | 1.01 (0.04) | 0.00 (-0.00, 0.00) |
| median [IQR] | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | - (-, -) | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | - (-, -) |
| min, max | 0.80, 1.67 | 0.80, 1.50 | - (-, -) | 0.80, 1.50 | 0.80, 1.50 | - (-, -) |
| <u> </u> | | • | | | | |

Appendix 7. Balance Assessment - Table 1

| Interest (1997) Propose From (1997) Prop | | | | | | | |
|---|---|---|---|---|---|---|---|
| March Marc | MARKETSCAN | | | | | | |
| March Marc | Variable | | | | | | |
| 2002 er 09 1412092001 1412092001 1412092001 141209001 14 | | 68,932 | 25,357 | - (-, -) | 25,346 | 25,346 | - (-, -) |
| 2002 1976 | | | | | | | |
| Section Sect | 7 7 7 | -, , | | | | | |
| SEARCH S | | 49,520 (71.8%) | 20,702 (81.6%) | -9.8% (-10.4%, -9.2%) | 20,846 (82.2%) | 20,692 (81.6%) | 0.6% (-0.1%, 1.3%) |
| | Age | | | | | | |
| 1800 5500 1800 5500 1800 5500 1800 5500 1800 5500 1800 5500 1800 5500 1500 5500 5 | | | | | | | |
| 1.23144279 | | | | ( ) / | | | |
| September 1,700 | | | | | | | |
| Nembeat Pri 19 229 (1879) 239 (1879) 2 | | 30,788 (44.7%) | 11,243 (44.3%) | 0.3% (-0.4%, 1.0%) | 11,307 (44.6%) | 11,240 (44.3%) | 0.3% (-0.6%, 1.1%) |
| Mayes Franciscont on (%) | | 7 701 (11 00() | 2102 (2.00) | 2.50/ /2.10/ 2.00/) | 2107 (0.70) | 2102 (0.70) | 0.00/ / 0.50/ 0.50/ |
| Sommor | | | | | | | |
| Medic 4 Miles | | | | | | | |
| Manage (19) | | | | | | | |
| Communication (19) | | | | | | | |
| Contempt | | | | | | | |
| Commentation Comm | | 6,749 (9.8%) | 2,319 (9.1%) | 0.6% (0.2%, 1.1%) | 2,305 (9.1%) | 2,318 (9.1%) | -0.1% (-0.6%, 0.5%) |
| Class 10 molesy m | | 2 242 /2 20/ | | | | | |
| Class 2 Oberlay, (196) | | | | | | | |
| Class 3 Dissip; (n 16) | | | | | | | |
| Unspectfold Design (19) | | | | | | | |
| 1.35 (6.529) 3.36 (6.529) 3.36 (6.529) 3.36 (6.529) 3.37 (6.529) 3.26 (2.129) 3.34 (1.250) 3.3 | | | | | | | |
| abetic nepropathy; (19) 3.34 (13.5%) 3.34 (13.5%) 3.34 (13.5%) 3.34 (13.5%) 3.34 (13.5%) 3.34 (13.5%) 3.34 (13.5%) 3.35 (10.9%) 3.37 (10.9%) 3.38 (10.9%) 3.38 (10.9%) 3.39 ( | | | | | | | |
| indect. experimentary, (%) aboles with other operiment in complications; (%) 94 (14%) 39 (13%) 29 (14%) 39 (13%) 39 (14%) 39 (13%) 39 (14%) 39 (13%) 39 (14%) 39 (13%) 39 (14%) 39 (14%) 39 (13%) 39 (14%) 39 (14 | | | | | | | |
| alseles with order optivalnic complexations. in (%) 4,788 (6.9%) 4,788 (6.9%) 1,781 (6.9%) 4,781 (6.9%) 4,78 | | | | | | | |
| allestes with perinternal circulatory disorders; n (%) 976 (1.4%) | | | | | | | |
| labelet for, fi (%) 294 (4.8%) 326 (3.4%) 0.1% (0.0%, 6.3%) 37 (1.3%) 320 (1.3%) 0.0% (0.2%, 0.2%) 294 (3.6%) 82 (3.4%) 1.0% (1.5%) 894 (3.5%) 894 (3.5%) 81 (3.4%) 0.1% (0.2%, 6.5%) 294 (3.6%) 1.23 (4.85%) 1.23 (4.85%) 1.25 (4.83%) 1.22 | | | ( ) | | | 1 | |
| recitle dysheriors n (%) 1881 173% 1.600 (181%) 1.838 1173% 1.600 (181%) 1.838 1173% 1.600 (181%) 1.838 1173% 1.600 (181%) 1.838 1173% 1.8 | | | | | | | |
| 1,238,1172% 4,500 (18.1%) 1.0% (-1.5% -0.4%) 4,533 (17.9%) 4,594 (18.1%) -0.2% (-0.7% -0.4%) 4,533 (17.9%) 12.25 (-1.4.5%) -0.2% (-0.7% -0.4%) 4.533 (17.9%) 12.25 (-1.4.5%) -0.2% (-1.7% -0.3%) 12.25 (-1.4.5%) -0.2% (-1.7% -0.3%) 12.25 (-1.4.5%) -0.2% (-1.7% -0.3%) -0.2% (-1.2% -0.3%) -0.2% (- | | | | | | | |
| 229146.5% 129146.5% 1291 | | | | | | | |
| Initinetations.nr (%) | | | | | | | |
| Libile angins; n (%) 1.008 (1.5%) 2.80 (1.1%) 2.80 (1.1%) 3.0% (1.0%) 3.0% (1. | | | | | | | |
| Instable anginez, n (%) 288 (11%) 287 (11%) 288 (11%) 288 (11%) 287 (11%) 287 (11%) 287 (11%) 288 (11%) 288 (11%) 287 (11%) 287 (11%) 287 (11%) 288 (11%) 288 (11%) 287 (11%) 287 (11%) 288 (11%) 288 (11%) 287 (11%) 288 (11%) 288 (11%) 287 (11%) 288 (11%) 288 (11%) 287 (11%) 287 (11%) 287 (11%) 288 (11%) 288 (11%) 287 (11%) 287 (11%) 287 (11%) 287 (11%) 288 (11%) 288 (11%) 287 (11%) 287 (11%) 288 (11%) 287 (11%) 288 (11%) 287 (11%) 287 (11%) 287 (11%) 288 (11%) 287 (11%) 288 (11%) 287 (11%) 288 (11%) 287 (11%) 288 (11%) 288 (11%) 287 (11%) 288 (11%) 288 (11%) 287 (11%) 287 (11%) 288 (11%) 288 (11%) 287 (11%) 287 (11%) 288 (11%) 288 (11%) 288 | | | | | | | |
| ypertnesiscn (1 (%) | | | | | | | |
| yperfunctering n (%) | | | | | | | |
| trial fibrillation: n (%) 3.32 fc (4.8%) 11.09 (4.4%) 0.5% (0.2%, 0.8%) 11.36 (4.5%) 11.09 (4.4%) 0.1% (-0.3%, 0.5%) revious cardiac conduction disorder: n (%) 1.885 (2.7%) 6.03 (2.4%) 0.4% (0.1%, 0.4%) 227 (0.9%) 229 (0.9%) 2.20 (0.9%) 229 (0.9%) 220 (0.9%) 230 (3.9%) 333 (3.9%) | | | | | | | |
| ardiac conduction disorder, n (%) 603 (2.4%) 608 (2.4%) 608 (2.4%) 609 (0.0% (0.3%, 0.3%) 808 (2.4%) 609 (0.0% (0.2%, 0.3%) 29 (0.9%) 609 (0.2% (0.1%, 0.4%) 27 (0.9%) 29 (0.9%) 608 (0.2% (0.2%) 608 (0.2% (0.1%, 0.4%) 608 (0.2% (0.1%, 0.4%) 608 (0.2% (0.1%, 0.2%) 608 (0.2% (0.1%, 0.4%) 608 (0.2% (0.1%) 608 (0.2% | | | | | | | |
| revious cardiac procedure (CABG, PTCA, Stent); n (%) | | | | | | | |
| Chemic stroke; n (%) | | | | | | | |
| VD diagnosis or surgery; n (%) 2,303 (3.3%) 9,532 (13.8%) | | | . , , | | | , | |
| ther cardiac dysrhythmia; n (%) 9,532 (13.8%) 9,532 (13.8%) 3,341 (13.2%) 0,7% (0.2%, 1.1%) 3,371 (13.3%) 3,339 (13.2%) 0,1% (0.5%, 0.7%) ardiomyopathy; n (%) 1,697 (2.8%) 598 (2.4%) 0,4% (0.2%, 0.6%) 576 (2.3%) 588 (2.4%) 0,1% (0.4%, 0.2%) 4.0% (0.4%, 0.2%) 588 (2.4%) 0,1% (0.4%, 0.2%) 4.0% (0.4%, 0.4%) 4.0% (0.5%, 0.1%) 4.0% (0.5%, 0.1%) 4.0% (0.3%) | | | | | | | |
| ardiomyopathy; n (%) also (1,58%) also (1,58 | | | | | | | |
| alve disorders; n(%) 3,831 (5.6%) 1,292 (5.1%) 0,5% (0.1%, 0.8%) 1,286 (5.1%) 1,292 (5.1%) 0,0% (-0.4%, 0.4%) alve replacement; n(%) 326 (0.5%) 85 (0.3%) 0,1% (0.0%, 0.2%) 80 (0.3%) 1,280 (3.3%) 227 (0.9%) 1,711 (0.9%) 227 (0.9%) 1,771 (7.0%) 1,771 (7 | | | | | | | |
| alve replacement; n (%) 326 (0.5%) 326 (0.5%) 327 (0.9%) 711 (1.0%) 712 (1.0%) 713 (1.0%) 714 (1.0%) 714 (1.0%) 714 (1.0%) 715 ( | Valve disorders; n (%) | | | | | | |
| IA; n (%) 711 (1.0%) 227 (0.9%) 0.1% (-0.0%, 0.3%) 214 (0.8%) 227 (0.9%) -0.1% (-0.2%, 0.1%) dema; n (%) 4.973 (7.2%) 1,771 (7.0%) 0.2% (-0.1%, 0.6%) 1,794 (7.1%) 1,771 (7.0%) 0.1% (-0.4%, 0.5%) enous thromboembolism; Pulmonary embolism; n (%) 1,483 (2.2%) 504 (2.0%) 0.2% (-0.0%, 0.4%) 486 (1.9%) 504 (2.0%) -0.1% (-0.3%, 0.2%) ulmonary hypertension; n (%) 754 (1.1%) 238 (0.9%) 0.2% (0.0%, 0.3%) 245 (1.0%) 238 (0.9%) 0.0% (-0.1%, 0.2%) mplantable cardioverter defibrillator; n (%) 115 (0.2%) 33 (0.1%) 0.0% (-0.0%, 0.1%) 39 (0.2%) 33 (0.1%) 0.0% (-0.0%, 0.1%) 288 (0.9%) 0.0% (-0.0%, 0.1%) 39 (0.2%) 33 (0.1%) 0.0% (-0.0%, 0.1%) 39 (0.2%) 33 (0.1%) 0.0% (-0.0%, 0.1%) 39 (0.2%) 33 (0.1%) 0.0% (-0.0%, 0.1%) 39 (0.2%) 33 (0.1%) 0.0% (-0.0%, 0.1%) 39 (0.2%) 33 (0.1%) 0.0% (-0.0%, 0.0%) 267 (1.1%) 251 (1.0%) 0.1% (-0.1%, 0.0%) 267 (1.1%) 251 (0.0%) 0.1% (-0.1%, 0.0%) 4.243 (9.6%) 2452 (9.7%) -1.0% (0.0%, 0.0%) 1.0% (0.0%) 0.0% (-0.0%, 0.0%) 9.0% 0.0% (-0.0%, 0.0%) | Valve replacement; n (%) | | | | | | |
| dema; n (%) 4,973 (7.2%) 1,771 (7.0%) 0.2% (-0.1%, 0.6%) 1,794 (7.1%) 1,771 (7.0%) 0.1% (-0.4%, 0.5%) enous thromboembolism; n (%) 1,483 (2.2%) 504 (2.0%) 0.2% (-0.0%, 0.4%) 486 (1.9%) 504 (2.0%) -0.1% (-0.3%, 0.2%) ulmonary hypertension; n (%) 754 (1.1%) 238 (0.9%) 0.2% (0.0%, 0.3%) 245 (1.0%) 238 (0.9%) 0.0% (-0.0%, 0.2%) nplantable cardioverter defibrillator; n (%) 115 (0.2%) 33 (0.1%) 0.0% (-0.0%, 0.1%) 39 (0.2%) 33 (0.1%) 0.0% (-0.0%, 0.1%) 39 (0.2%) 33 (0.1%) 0.0% (-0.0%, 0.1%) 39 (0.2%) 33 (0.1%) 0.0% (-0.0%, 0.1%) 39 (0.2%) 33 (0.1%) 0.0% (-0.0%, 0.1%) 39 (0.2%) | TIA; n (%) | | | | | | |
| enous thromboembolism / Pulmonary embolism; n (%) | Edema; n (%) | | | | | | |
| Implantable cardioverter defibrillator; n (%) 115 (0.2%) 33 (0.1%) 0.0% (-0.0%, 0.1%) 39 (0.2%) 33 (0.1%) 0.0% (-0.0%, 0.1%) yperkalemis; n (%) 887 (1.3%) 251 (1.0%) 0.3% (0.1%, 0.4%) 267 (1.1%) 251 (1.0%) 0.1% (-0.1%, 0.2%) oronary atherosclerosis; n (%) 7,620 (11.1%) 2,452 (9.7%) 1.44 (0.9%, 1.8%) 2,423 (9.6%) 2,452 (9.7%) -0.1% (-0.6%, 0.4%) erebrovascular procedure; n (%) 31 (0.0%) 9 (0.0%) 0.0% (-0.0%, 0.0%) 7 (0.0%) 9 (0.0%) -0.0% (-0.0%, 0.0%) KD stage 1-2; n (%) 29 (0.0%) 9 (0.0%) 0.0% (-0.0%, 0.0%) 8 (0.0%) 9 (0.0%) -0.0% (-0.0%, 0.0%) KD stage 3-4; n (%) 1,349 (2.0%) 521 (2.1%) -0.1% (-0.4%, 0.1%) 492 (1.9%) 521 (2.1%) -0.1% (-0.4%, 0.1%) KD stage 3-4; n (%) 1,206 (1.7%) 367 (1.4%) 0.3% (0.0%, 0.5%) 1,049 (4.1%) 1,069 (4.2%) -0.1% (-0.4%, 0.3%) nspecified CKD; n (%) 1,206 (1.7%) 367 (1.4%) 0.3% (0.0%, 0.5%) 381 (1.5%) 367 (1.4%) 0.1% (-0.4%, 0.3%) cute kidney injury; n (%) 1,823 | Venous thromboembolism / Pulmonary embolism; n (%) | 1,483 (2.2%) | 504 (2.0%) | 0.2% (-0.0%, 0.4%) | 486 (1.9%) | 504 (2.0%) | -0.1% (-0.3%, 0.2%) |
| Implantable cardioverter defibrillator; n (%) 115 (0.2%) 33 (0.1%) 0.0% (-0.0%, 0.1%) 39 (0.2%) 33 (0.1%) 0.0% (-0.0%, 0.1%) yperkalemis; n (%) 887 (1.3%) 251 (1.0%) 0.3% (0.1%, 0.4%) 267 (1.1%) 251 (1.0%) 0.1% (-0.1%, 0.2%) oronary atherosclerosis; n (%) 7,620 (11.1%) 2,452 (9.7%) 1.44 (0.9%, 1.8%) 2,423 (9.6%) 2,452 (9.7%) -0.1% (-0.6%, 0.4%) erebrovascular procedure; n (%) 31 (0.0%) 9 (0.0%) 0.0% (-0.0%, 0.0%) 7 (0.0%) 9 (0.0%) -0.0% (-0.0%, 0.0%) KD stage 1-2; n (%) 29 (0.0%) 9 (0.0%) 0.0% (-0.0%, 0.0%) 8 (0.0%) 9 (0.0%) -0.0% (-0.0%, 0.0%) KD stage 3-4; n (%) 1,349 (2.0%) 521 (2.1%) -0.1% (-0.4%, 0.1%) 492 (1.9%) 521 (2.1%) -0.1% (-0.4%, 0.1%) KD stage 3-4; n (%) 1,206 (1.7%) 367 (1.4%) 0.3% (0.0%, 0.5%) 1,049 (4.1%) 1,069 (4.2%) -0.1% (-0.4%, 0.3%) nspecified CKD; n (%) 1,206 (1.7%) 367 (1.4%) 0.3% (0.0%, 0.5%) 381 (1.5%) 367 (1.4%) 0.1% (-0.4%, 0.3%) cute kidney injury; n (%) 1,823 | Pulmonary hypertension; n (%) | 754 (1.1%) | 238 (0.9%) | 0.2% (0.0%, 0.3%) | 245 (1.0%) | 238 (0.9%) | 0.0% (-0.1%, 0.2%) |
| $ \begin{array}{c} \text{coronary atherosclerosis; n (\%)} & 7,620 (111\%) & 2,452 (9.7\%) & 1.4\% (0.9\%, 1.8\%) & 2,423 (9.6\%) & 2,452 (9.7\%) & -0.1\% (-0.6\%, 0.4\%) \\ \text{erebrovascular procedure; n (\%)} & 31 (0.0\%) & 9 (0.0\%) & 0.0\% (-0.0\%, 0.0\%) & 7 (0.0\%) & 9 (0.0\%) & -0.0\% (-0.0\%, 0.0\%) \\ \text{seption of pacemakers / removal of cardiac lead; n (\%)} & 13 (0.0\%) & 9 (0.0\%) & 0.0\% (-0.0\%, 0.0\%) & 8 (0.0\%) & 9 (0.0\%) & -0.0\% (-0.0\%, 0.0\%) \\ \text{KD stage 1-2; n (\%)} & 1,349 (2.0\%) & 521 (2.1\%) & -0.1\% (-0.3\%, 0.1\%) & 492 (1.9\%) & 521 (2.1\%) & -0.1\% (-0.4\%, 0.1\%) \\ \text{KD stage 3-4; n (\%)} & 3,386 (4.9\%) & 1.669 (4.2\%) & 0.7\% (0.4\%, 1.0\%) & 1.049 (4.1\%) & 1.069 (4.2\%) & -0.1\% (-0.4\%, 0.3\%) \\ \text{RD stage 3-4; n (\%)} & 3,386 (4.9\%) & 1.206 (1.7\%) & 367 (1.4\%) & 0.3\% (0.1\%, 0.5\%) & 381 (1.5\%) & 367 (1.4\%) & 0.1\% (-0.4\%, 0.3\%) \\ \text{cute kidney injury; n (\%)} & 1,823 (2.6\%) & 604 (2.4\%) & 0.3\% (0.0\%, 0.5\%) & 618 (2.4\%) & 604 (2.4\%) & 0.1\% (-0.2\%, 0.3\%) \\ \text{supertensive nephropathy; n (\%)} & 3,012 (4.4\%) & 1,039 (4.1\%) & 0.3\% (-0.0\%, 0.6\%) & 1,031 (4.1\%) & 1.039 (4.1\%) & 0.0\% (-0.4\%, 0.3\%) \\ \text{rinary tact infections; n (\%)} & 6,196 (9.0\%) & 2,374 (9.4\%) & 0.2\% (-0.8\%, 0.3\%) & 921 (3.9\%) & 925 (3.6\%) & 0.2\% (-0.4\%, 0.4\%) & 948 (3.7\%) & 925 (3.6\%) & 0.1\% (-0.2\%, 0.3\%) \\ \text{roll thiasis (Kidney and urinary stone); n (\%)} & 2,744 (4.0\%) & 1,007 (4.0\%) & 1,007 (4.0\%) & 991 (3.3\%) & 91 (3.07 (4.0\%) & -0.1\% (-0.2\%, 0.3\%) \\ \text{roll thiasis (Kidney and urinary stone); n (\%)} & 2,744 (4.0\%) & 1,007 (4.0\%) & 0.0\% (-0.3\%, 0.3\%) & 991 (3.9\%) & 1,007 (4.0\%) & -0.1\% (-0.2\%, 0.3\%) \\ \text{roll thiasis (Kidney and urinary stone); n (\%)} & 2,744 (4.0\%) & 1,007 (4.0\%) & 0.0\% (-0.3\%, 0.3\%) & 991 (3.9\%) & 1,007 (4.0\%) & -0.1\% (-0.4\%, 0.3\%) \\ \text{roll thiasis (Kidney and urinary stone); n (\%)} & 2,744 (4.0\%) & 1,007 (4.0\%) & 1,007 (4.0\%) & 0.0\% (-0.3\%, 0.3\%) & 991 (3.9\%) & 1,007 (4.0\%) & -0.1\% (-0.4\%, 0.3\%) \\ ro$ | Implantable cardioverter defibrillator, n (%) | 115 (0.2%) | 33 (0.1%) | 0.0% (-0.0%, 0.1%) | | 33 (0.1%) | 0.0% (-0.0%, 0.1%) |
| erebrovascular procedure; n (%) 31 (0.0%) 9 (0.0%) 0.0% (-0.0%, 0.0%) 7 (0.0%) 9 (0.0%) -0.0% (-0.0%, 0.0%) sertion of pacemakers / removal of cardiac lead; n (%) 29 (0.0%) 9 (0.0%) 0.0% (-0.0%, 0.0%) 8 (0.0%) 9 (0.0%) 9 (0.0%) -0.0% (-0.0%, 0.0%) 8 (0.0%) 9 (0.0%) 9 (0.0%) -0.0% (-0.0%, 0.0%) 8 (0.0%) 9 (0.0%) 9 (0.0%) -0.0% (-0.0%, 0.0%) 8 (0.0%) 9 (0.0%) 9 (0.0%) -0.0% (-0.0%, 0.0%) 8 (0.0%) 9 | Hyperkalemia; n (%) | 887 (1.3%) | 251 (1.0%) | 0.3% (0.1%, 0.4%) | 267 (1.1%) | 251 (1.0%) | 0.1% (-0.1%, 0.2%) |
| sertion of pacemakers / removal of cardiac lead; n (%) 29 (0.0%) 9 (0.0%) 0.0% (-0.0%, 0.0%) 8 (0.0%) 9 (0.0%) -0.0% (-0.0%, 0.0%) 8 (0.0%) 9 (0.0%) -0.0% (-0.0%, 0.0%) 8 (0.0%) 9 (0.0%) -0.0% (-0.0%, 0.0%) 9 (0.0%) -0.0% (-0.0%, 0.0%) 8 (0.0%) 9 (0.0%) -0.0% (-0.0%, 0.0%) 1349 (2.0%) 521 (2.1%) -0.1% (-0.4%, 0.1%) 10.09 (4.2%) -0.1% (-0.4%, 0.1%) 10.09 (4.1%) 10.09 (4.1%) 10.09 (4.2%) 10.09 (4.1%) 10.09 (4.1%) 10.09 (4.1%) 10.09 (4.1%) 10.09 (4.2%) 10.09 (4.1%) 10.09 | Coronary atherosclerosis; n (%) | 7,620 (11.1%) | 2,452 (9.7%) | 1.4% (0.9%, 1.8%) | 2,423 (9.6%) | 2,452 (9.7%) | -0.1% (-0.6%, 0.4%) |
| KD stage 1-2; n (%) | Cerebrovascular procedure; n (%) | 31 (0.0%) | | 0.0% (-0.0%, 0.0%) | 7 (0.0%) | 9 (0.0%) | -0.0% (-0.0%, 0.0%) |
| KD stage 3-4; n (%) | Insertion of pacemakers / removal of cardiac lead; n (%) | 29 (0.0%) | 9 (0.0%) | 0.0% (-0.0%, 0.0%) | 8 (0.0%) | 9 (0.0%) | -0.0% (-0.0%, 0.0%) |
| nspecified CKD; n (%) 1,206 (1.7%) 367 (1.4%) 0.3% (0.1%, 0.5%) 381 (1.5%) 367 (1.4%) 0.1% (-0.2%, 0.3%) cute kidney injury; n (%) 1,823 (2.6%) 604 (2.4%) 0.3% (0.0%, 0.5%) 618 (2.4%) 604 (2.4%) 0.1% (-0.2%, 0.3%) ypertensive nephropathy; n (%) 3,012 (4.4%) 1,039 (4.1%) 0.3% (-0.0%, 0.6%) 1,031 (4.1%) 1,039 (4.1%) -0.0% (-0.4%, 0.3%) initiary tract infections; n (%) 6,196 (9.0%) 2,374 (9.4%) -0.4% (-0.8%, 0.0%) 2,397 (9.5%) 2,372 (9.4%) -0.1% (-0.4%, 0.6%) enital infections; n (%) 2,619 (3.8%) 925 (3.6%) 0.2% (-0.1%, 0.4%) 948 (3.7%) 925 (3.6%) 0.1% (-0.2%, 0.3%) rolithiasis (Kidney and urinary stone); n (%) 2,744 (4.0%) 1,007 (4.0%) 0.0% (-0.3%, 0.3%) 991 (3.9%) 1,007 (4.0%) -0.1% (-0.4%, 0.3%) | CKD stage 1-2; n (%) | | | | | | |
| cute kidney injury; $n$ (%) 1,823 (2.6%) 604 (2.4%) 0.3% (0.0%, 0.5%) 618 (2.4%) 604 (2.4%) 0.1% (-0.2%, 0.3%) ypertensive nephropathy; $n$ (%) 3,012 (4.4%) 1,039 (4.1%) 0.3% (-0.0%, 0.6%) 1,031 (4.1%) 1,039 (4.1%) -0.0% (-0.4%, 0.3%) rinary tract infections; $n$ (%) 6,196 (9.0%) 2,374 (9.4%) -0.4% (-0.8%, 0.0%) 2,397 (9.5%) 2,372 (9.4%) 0.1% (-0.4%, 0.6%) enital infections; $n$ (%) 2,619 (3.8%) 925 (3.6%) 0.2% (-0.1%, 0.4%) 948 (3.7%) 925 (3.6%) 0.1% (-0.2%, 0.4%) rolithiasis (Kidney and urinary stone); $n$ (%) 2,744 (4.0%) 1,007 (4.0%) 0.0% (-0.3%, 0.3%) 991 (3.9%) 1,007 (4.0%) -0.1% (-0.4%, 0.3%) | CKD stage 3-4; n (%) | | | | | | |
| $ ypertensive nephropathy; n (\%) \\ 3,012 (4.4\%) \\ 5,196 (9.0\%) \\ 2,374 (9.4\%) \\ 2,619 (3.8\%) \\ 925 (3.6\%) \\ 1,039 (4.1\%) \\ 2,04 (9.0\%, 0.6\%) \\ 2,374 (9.4\%) \\ 2,274 (4.0\%) \\ 2,274 (4.0\%)$ | Unspecified CKD; n (%) | | | | | | |
| $\begin{array}{cccccccccccccccccccccccccccccccccccc$ | Acute kidney injury; n (%) | 1,823 (2.6%) | 604 (2.4%) | 0.3% (0.0%, 0.5%) | 618 (2.4%) | 604 (2.4%) | 0.1% (-0.2%, 0.3%) |
| enital infections; n (%) 2.619 (3.8%) 925 (3.6%) 0.2% (-0.1%, 0.4%) 948 (3.7%) 925 (3.6%) 0.1% (-0.2%, 0.4%) rolithiasis (Kidney and urinary stone); n (%) 2,744 (4.0%) 1,007 (4.0%) 0.0% (-0.3%, 0.3%) 991 (3.9%) 1,007 (4.0%) -0.1% (-0.4%, 0.3%) | Hypertensive nephropathy; n (%) | 3,012 (4.4%) | | | | | -0.0% (-0.4%, 0.3%) |
| rolithiasis (Kidney and urinary stone); $n$ (%) 2,744 (4.0%) 1,007 (4.0%) 0.0% (-0.3%, 0.3%) 991 (3.9%) 1,007 (4.0%) -0.1% (-0.4%, 0.3%) | Urinary tract infections; n (%) | | | | | | |
| | Genital infections; n (%) | 2,619 (3.8%) | 925 (3.6%) | | | | |
| $\begin{array}{cccccccccccccccccccccccccccccccccccc$ | Urolithiasis (Kidney and urinary stone); n (%) | | | | | | |
| | COPD; n (%) | 2,880 (4.2%) | 930 (3.7%) | 0.5% (0.2%, 0.8%) | 939 (3.7%) | 930 (3.7%) | 0.0% (-0.3%, 0.4%) |

| | | 1 | 1 | Ī | 1 | 1 |
|---|---|---|---|---|---|---|
| Asthma; n (%) | 6,552 (9.5%) | 2,362 (9.3%) | 0.2% (-0.2%, 0.6%) | 2,394 (9.4%) | 2,361 (9.3%) | 0.1% (-0.4%, 0.6%) |
| Obstructive sleep apnea; n (%) | 20,051 (29.1%) | 7,581 (29.9%) | -0.8% (-1.5%, -0.1%) | 7,552 (29.8%) | 7,576 (29.9%) | -0.1% (-0.9%, 0.7%) |
| Serious bacterial infections; n (%) | 1,540 (2.2%) | 523 (2.1%) | 0.2% (-0.0%, 0.4%) | 527 (2.1%) | 523 (2.1%) | 0.0% (-0.2%, 0.3%) |
| Pneumonia; n (%) | 1,953 (2.8%) | 645 (2.5%) | 0.3% (0.1%, 0.5%) | 683 (2.7%) | 645 (2.5%) | 0.1% (-0.1%, 0.4%) |
| Liver disease; n (%) | 9,460 (13.7%) | 3,508 (13.8%) | -0.1% (-0.6%, 0.4%) | 3,545 (14.0%) | 3,505 (13.8%) | 0.2% (-0.4%, 0.8%) |
| MASH/MASLD; n (%) | 6,419 (9.3%) | 2,373 (9.4%) | -0.0% (-0.5%, 0.4%) | 2,405 (9.5%) | 2,371 (9.4%) | 0.1% (-0.4%, 0.6%) |
| Fractures / Falls; n (%) | 2,051 (3.0%) | 714 (2.8%) | 0.2% (-0.1%, 0.4%) | 744 (2.9%) | 714 (2.8%) | 0.1% (-0.2%, 0.4%) |
| Osteoporosis; n (%) | 879 (1.3%) | 289 (1.1%) | 0.1% (-0.0%, 0.3%) | 285 (1.1%) | 289 (1.1%) | -0.0% (-0.2%, 0.2%) |
| Osteoarthritis; n (%) | 13,474 (19.5%) | 4,815 (19.0%) | 0.6% (-0.0%, 1.1%) | 4,830 (19.1%) | 4,812 (19.0%) | 0.1% (-0.6%, 0.8%) |
| Depression; n (%) | 11,039 (16.0%) | 3,957 (15.6%) | 0.4% (-0.1%, 0.9%) | 4,009 (15.8%) | 3,955 (15.6%) | 0.2% (-0.4%, 0.9%) |
| Dementia; n (%) | 587 (0.9%) | 153 (0.6%) | 0.2% (0.1%, 0.4%) | 149 (0.6%) | 153 (0.6%) | -0.0% (-0.2%, 0.1%) |
| Delirium or psychosis; n (%) | 380 (0.6%) | 94 (0.4%) | 0.2% (0.1%, 0.3%) | 103 (0.4%) | 93 (0.4%) | 0.0% (-0.1%, 0.2%) |
| Anxiety; n (%) | 14,298 (20.7%) | 5,316 (21.0%) | -0.2% (-0.8%, 0.4%) | 5,303 (20.9%) | 5,313 (21.0%) | -0.0% (-0.8%, 0.7%) |
| Sleep disorders; n (%) | 16,638 (24.1%) | 6,375 (25.1%) | -1.0% (-1.6%, -0.4%) | 6,407 (25.3%) | 6,368 (25.1%) | 0.2% (-0.6%, 0.9%) |
| | | 3,494 (13.8%) | -0.1% (-0.6%, 0.4%) | 3,441 (13.6%) | 3,491 (13.8%) | -0.2% (-0.8%, 0.4%) |
| Anemia; n (%) | 9,429 (13.7%)<br>1.387 (2.0%) | | | | | |
| Influenza; n (%) | | 641 (2.5%) | -0.5% (-0.7%, -0.3%) | 656 (2.6%) | 640 (2.5%) | 0.1% (-0.2%, 0.3%) |
| COVID; n (%) | 9,821 (14.2%) | 3,324 (13.1%) | 1.1% (0.6%, 1.6%) | 3,335 (13.2%) | 3,323 (13.1%) | 0.0% (-0.5%, 0.6%) |
| Hyperthyroidism and other thyroid gland disorders; n (%) | 14,374 (20.9%) | 5,634 (22.2%) | -1.4% (-2.0%, -0.8%) | 5,644 (22.3%) | 5,629 (22.2%) | 0.1% (-0.7%, 0.8%) |
| Hypothyroidism; n (%) | 11,121 (16.1%) | 4,388 (17.3%) | -1.2% (-1.7%, -0.6%) | 4,408 (17.4%) | 4,384 (17.3%) | 0.1% (-0.6%, 0.8%) |
| Nephrotic syndrome; n (%) | 38 (0.1%) | 9 (0.0%) | 0.0% (-0.0%, 0.1%) | 10 (0.0%) | 9 (0.0%) | 0.0% (-0.0%, 0.0%) |
| Urinary incontinence; n (%) | 1,876 (2.7%) | 651 (2.6%) | 0.2% (-0.1%, 0.4%) | 635 (2.5%) | 650 (2.6%) | -0.1% (-0.3%, 0.2%) |
| Biliary disease; n (%) | 153 (0.2%) | 60 (0.2%) | -0.0% (-0.1%, 0.1%) | 56 (0.2%) | 60 (0.2%) | -0.0% (-0.1%, 0.1%) |
| Pancreatitis; n (%) | 74 (0.1%) | 27 (0.1%) | 0.0% (-0.0%, 0.0%) | 33 (0.1%) | 27 (0.1%) | 0.0% (-0.0%, 0.1%) |
| Bowel obstruction; n (%) | 88 (0.1%) | 34 (0.1%) | -0.0% (-0.1%, 0.0%) | 32 (0.1%) | 34 (0.1%) | -0.0% (-0.1%, 0.1%) |
| Gastroparesis; n (%) | 325 (0.5%) | 137 (0.5%) | -0.1% (-0.2%, 0.0%) | 140 (0.6%) | 137 (0.5%) | 0.0% (-0.1%, 0.1%) |
| Number of antidiabetic drugs on CED | | | | , | | |
| mean (sd) | 2.07 (0.97) | 2.06 (0.98) | 0.02 (0.00, 0.03) | 2.05 (0.98) | 2.06 (0.98) | -0.01 (-0.03, 0.01) |
| median [IQR] | 2.00 [1.00, 3.00] | 2.00 [1.00, 3.00] | - () | 2.00 [1.00, 3.00] | 2.00 [1.00, 3.00] | - () |
| min, max | 1.00. 7.00 | 1.00, 7.00 | - (-, -) | 1.00, 7.00 | 1.00, 7.00 | - (-, -) |
| | 36,250 (52.6%) | 12,709 (50.1%) | 2.5% (1.7%, 3.2%) | 12,637 (49.9%) | 12,706 (50.1%) | -0.3% (-1.1%, 0.6%) |
| Concomitant use or initiation of Metformin; n (%) | | | | | | |
| Concomitant use or initiation of Insulins; n (%) | 9,131 (13.2%) | 3,420 (13.5%) | -0.2% (-0.7%, 0.3%) | 3,395 (13.4%) | 3,418 (13.5%) | -0.1% (-0.7%, 0.5%) |
| Concomitant use or initiation of Sulfonylureas; n (%) | 9,014 (13.1%) | 2,805 (11.1%) | 2.0% (1.6%, 2.5%) | 2,803 (11.1%) | 2,805 (11.1%) | -0.0% (-0.6%, 0.5%) |
| Concomitant use or initiation of DPP-4i; n (%) | 4,614 (6.7%) | 1,630 (6.4%) | 0.3% (-0.1%, 0.6%) | 1,642 (6.5%) | 1,629 (6.4%) | 0.1% (-0.4%, 0.5%) |
| Concomitant use or initiation of SGLT-2i; n (%) | 12,489 (18.1%) | 5,234 (20.6%) | -2.5% (-3.1%, -1.9%) | 5,085 (20.1%) | 5,228 (20.6%) | -0.6% (-1.3%, 0.1%) |
| Concomitant use or initiation of Any other glucose-lowering drugs; n (%) | 2,525 (3.7%) | 1,000 (3.9%) | -0.3% (-0.6%, -0.0%) | 998 (3.9%) | 1,000 (3.9%) | -0.0% (-0.4%, 0.3%) |
| Past use of Metformin; n (%) | 48,294 (70.1%) | 17,285 (68.2%) | 1.9% (1.2%, 2.6%) | 17,164 (67.7%) | 17,281 (68.2%) | -0.5% (-1.3%, 0.4%) |
| Past use of Insulins; n (%) | 12,548 (18.2%) | 4,794 (18.9%) | -0.7% (-1.3%, -0.1%) | 4,753 (18.8%) | 4,792 (18.9%) | -0.2% (-0.8%, 0.5%) |
| Past use of Sulfonylureas; n (%) | 12,888 (18.7%) | 4,197 (16.6%) | 2.1% (1.6%, 2.7%) | 4,238 (16.7%) | 4,197 (16.6%) | 0.2% (-0.5%, 0.8%) |
| Past use of DPP-4i; n (%) | 7,640 (11.1%) | 2,680 (10.6%) | 0.5% (0.1%, 1.0%) | 2,689 (10.6%) | 2,679 (10.6%) | 0.0% (-0.5%, 0.6%) |
| Past use of SGLT-2i; n (%) | 16,536 (24.0%) | 6,902 (27.2%) | -3.2% (-3.9%, -2.6%) | 6,748 (26.6%) | 6,895 (27.2%) | -0.6% (-1.4%, 0.2%) |
| Past use of Any other glucose-lowering drugs; n (%) | 3,705 (5.4%) | 1,450 (5.7%) | -0.3% (-0.7%, -0.0%) | 1,427 (5.6%) | 1,449 (5.7%) | -0.1% (-0.5%, 0.3%) |
| ACE-is/ARB's; n (%) | 47,681 (69.2%) | 17,598 (69.4%) | -0.2% (-0.9%, 0.4%) | 17,545 (69.2%) | 17,590 (69.4%) | -0.2% (-1.0%, 0.6%) |
| ARNI; n (%) | 873 (1.3%) | 291 (1.1%) | 0.1% (-0.0%, 0.3%) | 295 (1.2%) | 290 (1.1%) | 0.0% (-0.2%, 0.2%) |
| Thiazides; n (%) | 24,036 (34.9%) | 8,888 (35.1%) | -0.2% (-0.9%, 0.5%) | 8,847 (34.9%) | 8,884 (35.1%) | -0.1% (-1.0%, 0.7%) |
| Beta-blockers; n (%) | 22,154 (32.1%) | 7,988 (31.5%) | 0.6% (-0.0%, 1.3%) | 7,981 (31.5%) | 7,983 (31.5%) | -0.1% (-1.0%, 0.7%) |
| Calcium channel blockers; n (%) | 19,450 (28.2%) | 6,861 (27.1%) | 1.2% (0.5%, 1.8%) | 6,799 (26.8%) | 6,859 (27.1%) | -0.2% (-1.0%, 0.5%) |
| Digoxin / Digitoxin; n (%) | 205 (0.3%) | 75 (0.3%) | 0.0% (-0.1%, 0.1%) | 76 (0.3%) | 75 (0.3%) | 0.0% (-0.1%, 0.1%) |
| Loop diuretics; n (%) | 6,619 (9.6%) | 2,283 (9.0%) | 0.6% (0.2%, 1.0%) | 2,247 (8.9%) | 2,282 (9.0%) | -0.1% (-0.6%, 0.4%) |
| Other diuretics; n (%) | 5,294 (7.7%) | 1,887 (7.4%) | 0.2% (-0.1%, 0.6%) | 1,899 (7.5%) | 1,885 (7.4%) | 0.1% (-0.4%, 0.5%) |
| Intravenous diuretics; n (%) | 421 (0.6%) | 119 (0.5%) | 0.1% (0.0%, 0.2%) | 117 (0.5%) | 119 (0.5%) | -0.0% (-0.1%, 0.1%) |
| Nitrates; n (%) | 2,462 (3.6%) | 766 (3.0%) | 0.6% (0.3%, 0.8%) | 775 (3.1%) | 766 (3.0%) | 0.0% (-0.3%, 0.3%) |
| Anti-arrhythmics; n (%) | 989 (1.4%) | 333 (1.3%) | 0.1% (-0.0%, 0.3%) | 334 (1.3%) | 333 (1.3%) | 0.0% (-0.2%, 0.2%) |
| Statins; n (%) | 50,078 (72.6%) | 17,918 (70.7%) | 2.0% (1.3%, 2.6%) | 17,838 (70.4%) | 17,910 (70.7%) | -0.3% (-1.1%, 0.5%) |
| PCSK9 inhibitors and other lipid-lowering drugs; n (%) | 8,074 (11.7%) | 3,030 (11.9%) | -0.2% (-0.7%, 0.2%) | 3,062 (12.1%) | 3,028 (11.9%) | 0.1% (-0.4%, 0.7%) |
| Antiplatelet medications; n (%) | 5,332 (7.7%) | 1,767 (7.0%) | 0.8% (0.4%, 1.1%) | 1,704 (6.7%) | 1,766 (7.0%) | -0.2% (-0.7%, 0.2%) |
| Oral anticoagulants; n (%) | 4,225 (6.1%) | 1,461 (5.8%) | 0.4% (0.0%, 0.7%) | 1,492 (5.9%) | 1,461 (5.8%) | 0.1% (-0.3%, 0.5%) |
| COPD/Asthma medications; n (%) | 22,894 (33.2%) | 8,474 (33.4%) | -0.2% (-0.9%, 0.5%) | 8,525 (33.6%) | 8,467 (33.4%) | 0.2% (-0.6%, 1.1%) |
| NSAIDS: n (%) | 23,869 (34.6%) | 8,929 (35,2%) | -0.6% (-1.3%, 0.1%) | 8.926 (35.2%) | 8,923 (35.2%) | 0.0% (-0.8%, 0.8%) |
| Oral corticosteroids; n (%) | 19,020 (27.6%) | 7,236 (28.5%) | -0.9% (-1.6%, -0.3%) | 7,295 (28.8%) | 7,232 (28.5%) | 0.2% (-0.5%, 1.0%) |
| Osteoporosis agents (incl. bisphosphonates); n (%) | 903 (1.3%) | 329 (1.3%) | 0.0% (-0.2%, 0.2%) | 320 (1.3%) | 329 (1.3%) | -0.0% (-0.2%, 0.2%) |
| | 17,125 (24.8%) | 6,394 (25.2%) | -0.4% (-1.0%, 0.3%) | 6,423 (25.3%) | 6,389 (25.2%) | 0.1% (-0.6%, 0.9%) |
| Opioids; n (%) | | | | | | |
| Anti-depressants; n (%) | 24,872 (36.1%) | 9,373 (37.0%) | -0.9% (-1.6%, -0.2%) | 9,423 (37.2%) | 9,368 (37.0%) | 0.2% (-0.6%, 1.1%) |
| | | | 0.1% (-0.2%, 0.3%) | 754 (3.0%) | 754 (3.0%) | 0.0% (-0.3%, 0.3%) |
| Antipsychotics; n (%) | 2,092 (3.0%) | 755 (3.0%) | | | | |
| Anxiolytics / hypnotics, benzos; n (%) | 13,643 (19.8%) | 5,358 (21.1%) | -1.3% (-1.9%, -0.8%) | 5,347 (21.1%) | 5,352 (21.1%) | -0.0% (-0.7%, 0.7%) |
| | | | | | | -0.0% (-0.7%, 0.7%)<br>-0.0% (-0.1%, 0.1%) |
| Anxiolytics / hypnotics, benzos; n (%) | 13,643 (19.8%) | 5,358 (21.1%) | -1.3% (-1.9%, -0.8%) | 5,347 (21.1%) | 5,352 (21.1%) | |

| D | 1 | 1 | T | | T | 1 |
|---|---|---|---|---|---|---|
| Number of distinct medications | 12.01 (6.42) | 10.40 (0.50) | 0.07 / 0.00 0.10 | 12.46.46.60 | 12.40 (0.50) | 0.01 / 0.10 0.10 |
| mean (sd) | 13.21 (6.43)<br>12.00 [9.00, 17.00] | 13.48 (6.58)<br>12.00 [9.00, 17.00] | -0.27 (-0.36, -0.18)<br>- (-, -) | 13.46 (6.62)<br>12.00 [9.00, 17.00] | 13.48 (6.58)<br>12.00 [9.00, 17.00] | -0.01 (-0.13, 0.10)<br>- (-, -) |
| | 1.00, 72.00 | 1.00, 62.00 | | 1.00, 72.00 | 1.00, 62.00 | |
| min, max Number of office visits | 1.00, 72.00 | 1.00, 62.00 | - (-, -) | 1.00, 72.00 | 1.00, 62.00 | - (-, -) |
| mean (sd) | 8.35 (6.32) | 8.35 (6.21) | -0.00 (-0.09, 0.09) | 8.35 (6.33) | 8.35 (6.20) | 0.00 (-0.11, 0.11) |
| median [IQR] | 7.00 [4.00, 11.00] | 7.00 [4.00, 11.00] | - (-, -) | 7.00 [4.00, 11.00] | 7.00 [4.00, 11.00] | - (-, -) |
| min, max | 0.00, 107.00 | 0.00, 101.00 | - (-, -) | 0.00, 96.00 | 0.00, 101.00 | - (-, -) |
| Number of endocrinologist visits | 0.00, 107.00 | 0.00, 101.00 | - (-, -) | 0.00, 96.00 | 0.00, 101.00 | - (-, -) |
| mean (sd) | 0.33 (1.14) | 0.39 (1.24) | -0.06 (-0.07, -0.04) | 0.38 (1.30) | 0.39 (1.24) | -0.00 (-0.02, 0.02) |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - () |
| min, max | 0.00, 51.00 | 0.00, 63.00 | - (-, -) | 0.00, 51.00 | 0.00, 63.00 | - (-, -) |
| Number of cardiologist visits | 0.00, 3100 | 0.00, 03.00 | - (-, -) | 0.00, 31.00 | 0.00, 03.00 | - (-, -) |
| mean (sd) | 0.92 (2.53) | 0.83 (2.20) | 0.09 (0.06, 0.12) | 0.83 (2.41) | 0.83 (2.20) | -0.00 (-0.04, 0.04) |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | - (-, -) | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | - (-, -) |
| min, max | 0.00, 85.00 | 0.00, 49.00 | - (-, -) | 0.00, 80.00 | 0.00, 49.00 | - (-, -) |
| Number of internal/family medicine visits | 0.00, 03.00 | 0.00, 45.00 | (, ) | 0.00, 00.00 | 0.00, 45.00 | (7,7) |
| mean (sd) | 4.57 (5.14) | 4.55 (5.45) | 0.02 (-0.06, 0.10) | 4.55 (5.20) | 4.55 (5.45) | -0.00 (-0.10, 0.09) |
| median [IQR] | 3.00 [1.00, 6.00] | 3.00 [1.00, 6.00] | - (-, -) | 3.00 [1.00, 6.00] | 3.00 [1.00, 6.00] | - (-, -) |
| min, max | 0.00, 178.00 | 0.00, 364.00 | - (-, -) | 0.00, 178.00 | 0.00, 364.00 | - (-, -) |
| Number of Electrocardiograms (ECG/EKG) | 1.11,1,0.00 | | 111 | 2.2,2,0.00 | | 111 |
| mean (sd) | 0.73 (1.37) | 0.66 (1.23) | 0.07 (0.05, 0.09) | 0.66 (1.24) | 0.66 (1.23) | 0.01 (-0.02, 0.03) |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | -(-, -) | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | -() |
| min, max | 0.00, 35.00 | 0.00, 24.00 | - (-, -)<br>- (-, -) | 0.00, 35.00 | 0.00, 24.00 | - (-, -)<br>- (-, -) |
| Number of Echocardiograms | 5.55, 55.55 | 5.55, 27.00 | 117 | 5.55, 55.55 | 0.00, 24.00 | 10.7 |
| mean (sd) | 0.21 (0.62) | 0.19 (0.55) | 0.02 (0.02, 0.03) | 0.19 (0.57) | 0.19 (0.55) | -0.00 (-0.01, 0.01) |
| median (IOR) | 0.00 [0.00, 0.00] | 0.19 (0.55) | - (-, -) | 0.00 [0.00, 0.00] | 0.19 (0.03) | - (-, -) |
| min. max | 0.00, 22.00 | 0.00 [0.00, 0.00] | - (-, -) | 0.00.14.00 | 0.00, 11.00 | - (-, -) |
| Out-of-pocket medication cost | 0.00, 22.00 | 0.00, 11.00 | - (-, -) | 0.00, 14.00 | 0.00, 11.00 | - (-, -) |
| mean (sd) | 492.30 (905.36) | 561.98 (1,041.69) | -69.67 (-84.17, -55.18) | 540.98 (989.55) | 555.98 (912.47) | -15.00 (-31.57, 1.58) |
| median [IQR] | 287.51 [108.25, 618.62] | 311.20 [114.12, 701.32] | | 304.88 [112.98, 663.70] | 310.86 [114.07, 700.00] | -(-, -) |
| min, max | -31,469.49, 62,075.17 | -5,760.00, 54,171.99 | - (-, -)<br>- (-, -) | -19,471.05, 28,184.79 | -5,760.00, 32,501.25 | - (-, -)<br>- (-, -) |
| min, max Unique brand medicines | -31,469.49, 62,075.17 | -5,760.00, 54,171.99 | - (-, -) | -19,471.05, 28,184.79 | -5,760.00, 32,501.25 | - (-, -) |
| mean (sd) | 13.47 (6.61) | 13.70 (6.76) | -0.24 (-0.33, -0.14) | 13.68 (6.78) | 13.70 (6.75) | -0.02 (-0.14, 0.10) |
| median [IQR] | 12.00 [9.00, 17.00] | 12.00 [9.00, 17.00] | -(-, -) | 13.00 [9.00, 17.00] | 12.00 [9.00, 17.00] | - (-, -) |
| min, max | 1.00, 74.00 | 1.00, 62.00 | - (-, -)<br>- (-, -) | 1.00, 74.00 | 1.00, 62.00 | - (-, -)<br>- (-, -) |
| Unique generic medicines | 1.00, 74.00 | 1.00, 02.00 | - (-, -) | 1.00, 74.00 | 1.00, 02.00 | - (-, -) |
| mean (sd) | 13.21 (6.43) | 13.48 (6.58) | -0.27 (-0.36, -0.18) | 13.46 (6.62) | 13.48 (6.58) | -0.01 (-0.13, 0.10) |
| median [IQR] | 12.00 [9.00, 17.00] | 12.00 [9.00, 17.00] | -(-, -) | 12.00 [9.00, 17.00] | 12.00 [9.00, 17.00] | - (-, -) |
| min, max | 1.00, 72.00 | 1.00, 62.00 | - (-, -)<br>- (-, -) | 1.00, 72.00 | 1.00, 62.00 | - (-, -)<br>- (-, -) |
| Colonoscopy Sigmoidoscopy; n (%) | 7.654 (11.1%) | 2.748 (10.8%) | 0.3% (-0.2%, 0.7%) | 2.731 (10.8%) | 2.745 (10.8%) | -0.1% (-0.6%, 0.5%) |
| Flu Pneumococcal vaccine; n (%) | 19,111 (27.7%) | 6,589 (26.0%) | 1.7% (1.1%, 2.4%) | 6,635 (26.2%) | 6,586 (26.0%) | 0.2% (-0.6%, 0.3%) |
| Pap smear; n (%) | 8,443 (12.2%) | 3,301 (13.0%) | 1.7 70 (1.170, 2.44 70) | 0,033 (20.270) | | 0.2% (-0.6%, 1.0%) |
| PSA test; n (%) | | | 0.9% / 1.3% 0.3%) | 3 215 (12 7%) | | 0.3% ( 0.0% 0.3%) |
| | | | -0.8% (-1.3%, -0.3%) | 3,215 (12.7%) | 3,296 (13.0%) | -0.3% (-0.9%, 0.3%) |
| | 14,120 (20.5%) | 5,280 (20.8%) | -0.3% (-0.9%, 0.2%) | 5,355 (21.1%) | 3,296 (13.0%)<br>5,280 (20.8%) | 0.3% (-0.4%, 1.0%) |
| Fecal occult blood test; n (%) | 14,120 (20.5%)<br>2,496 (3.6%) | 5,280 (20.8%)<br>867 (3.4%) | -0.3% (-0.9%, 0.2%)<br>0.2% (-0.1%, 0.5%) | 5,355 (21.1%)<br>840 (3.3%) | 3,296 (13.0%)<br>5,280 (20.8%)<br>867 (3.4%) | 0.3% (-0.4%, 1.0%) -0.1% (-0.4%, 0.2%) |
| Fecal occult blood test; n (%) Bone mineral density tests; n (%) | 14,120 (20.5%)<br>2,496 (3.6%)<br>2,335 (3.4%) | 5,280 (20.8%)<br>867 (3.4%)<br>865 (3.4%) | -0.3% (-0.9%, 0.2%)<br>0.2% (-0.1%, 0.5%)<br>-0.0% (-0.3%, 0.2%) | 5,355 (21.1%)<br>840 (3.3%)<br>854 (3.4%) | 3,296 (13.0%)<br>5,280 (20.8%)<br>867 (3.4%)<br>865 (3.4%) | 0.3% (-0.4%, 1.0%)<br>-0.1% (-0.4%, 0.2%)<br>-0.0% (-0.4%, 0.3%) |
| Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) | 14,120 (20.5%)<br>2,496 (3.6%)<br>2,335 (3.4%)<br>18,887 (27.4%) | 5,280 (20.8%)<br>867 (3.4%)<br>865 (3.4%)<br>6,996 (27.6%) | -0.3% (-0.9%, 0.2%)<br>0.2% (-0.1%, 0.5%)<br>-0.0% (-0.3%, 0.2%)<br>-0.2% (-0.8%, 0.5%) | 5,355 (21.1%)<br>840 (3.3%)<br>854 (3.4%)<br>6,963 (27.5%) | 3,296 (13.0%)<br>5,280 (20.8%)<br>867 (3.4%)<br>865 (3.4%)<br>6,993 (27.6%) | 0.3% (-0.4%, 1.0%)<br>-0.1% (-0.4%, 0.2%)<br>-0.0% (-0.4%, 0.3%)<br>-0.1% (-0.9%, 0.7%) |
| Fecal occult blood test n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) | 14,120 (20.5%)<br>2,496 (3.6%)<br>2,335 (3.4%) | 5,280 (20.8%)<br>867 (3.4%)<br>865 (3.4%) | -0.3% (-0.9%, 0.2%)<br>0.2% (-0.1%, 0.5%)<br>-0.0% (-0.3%, 0.2%) | 5,355 (21.1%)<br>840 (3.3%)<br>854 (3.4%) | 3,296 (13.0%)<br>5,280 (20.8%)<br>867 (3.4%)<br>865 (3.4%) | 0.3% (-0.4%, 1.0%)<br>-0.1% (-0.4%, 0.2%)<br>-0.0% (-0.4%, 0.3%) |
| Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbA1C tests | 14,120 (20.5%)<br>2,496 (3.6%)<br>2,335 (3.4%)<br>18,887 (27.4%)<br>22,031 (32.0%) | 5,280 (20.8%)<br>867 (3.4%)<br>865 (3.4%)<br>6,996 (27.6%)<br>7,446 (29.4%) | -0.3% (-0.9%, 0.2%)<br>0.2% (-0.1%, 0.5%)<br>-0.0% (-0.3%, 0.2%)<br>-0.2% (-0.8%, 0.5%)<br>2.6% (1.9%, 3.3%) | 5,355 (21.1%)<br>840 (3.3%)<br>854 (3.4%)<br>6,963 (27.5%)<br>7,498 (29.6%) | 3,296 (13.0%)<br>5,280 (20.8%)<br>867 (3.4%)<br>865 (3.4%)<br>6,993 (27.6%)<br>7,442 (29.4%) | 0.3% (-0.4%, 1.0%)<br>-0.1% (-0.4%, 0.2%)<br>-0.0% (-0.4%, 0.3%)<br>-0.1% (-0.9%, 0.7%)<br>0.2% (-0.6%, 1.0%) |
| Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbAIC tests mean (sd) | 14,120 (20.5%)<br>2,496 (3.6%)<br>2,335 (3.4%)<br>18,887 (27.4%)<br>22,031 (32.0%)<br>213 (1.47) | 5,280 (20.8%)<br>867 (3.4%)<br>865 (3.4%)<br>6,996 (27.6%)<br>7,446 (29.4%)<br>2.18 (1.43) | -0.3% (-0.9%, 0.2%)<br>0.2% (-0.1%, 0.5%)<br>-0.0% (-0.3%, 0.2%)<br>-0.2% (-0.8%, 0.5%)<br>2.6% (1.9%, 3.3%)<br>-0.05 (-0.07, -0.03) | 5,355 (21.1%)<br>840 (3.3%)<br>854 (3.4%)<br>6,963 (27.5%)<br>7,498 (29.6%) | 3,296 (13.0%)<br>5,280 (20.8%)<br>867 (3.4%)<br>865 (3.4%)<br>6,993 (27.6%)<br>7,442 (29.4%) | 0.3% (-0.4%, 1.0%)<br>-0.1% (-0.4%, 0.2%)<br>-0.0% (-0.4%, 0.3%)<br>-0.1% (-0.9%, 0.7%)<br>0.2% (-0.6%, 1.0%)<br>-0.02 (-0.04, 0.01) |
| Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbA1C testsmean (sd)median [IQR] | 14,120 (20.5%)<br>2,496 (3.6%)<br>2,335 (3.4%)<br>18,887 (27.4%)<br>22,031 (32.0%)<br>213 (1.47)<br>200 (1.00, 3.00) | 5,280 (20.8%)<br>867 (3.4%)<br>865 (3.4%)<br>6,996 (27.6%)<br>7,446 (29.4%)<br>218 (1.43)<br>200 [1.00, 3.00] | -0.3% (-0.9%, 0.2%)<br>0.2% (-0.1%, 0.5%)<br>-0.0% (-0.3%, 0.2%)<br>-0.2% (-0.8%, 0.5%)<br>2.6% (1.9%, 3.3%)<br>-0.05 (-0.07, -0.03)<br>-(-,-) | 5,355 (21.1%)<br>840 (3.3%)<br>854 (3.4%)<br>6,963 (27.5%)<br>7,498 (29.6%)<br>217 (1.36)<br>2.00 [1.00, 3.00] | 3,296 (13.0%) 5,280 (20.8%) 867 (3.4%) 865 (3.4%) 6,993 (27.6%) 7,442 (29.4%) 218 (1.41) 2.00 [1.00, 3.00] | 0.3% (-0.4%, 1.0%)<br>-0.1% (-0.4%, 0.2%)<br>-0.0% (-0.4%, 0.3%)<br>-0.1% (-0.9%, 0.7%)<br>0.2% (-0.6%, 1.0%)<br>-0.02 (-0.04, 0.01)<br>-(-,-) |
| Fecal occult blood test n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbA1C testsmean (sd)median [IQR]min, max | 14,120 (20.5%)<br>2,496 (3.6%)<br>2,335 (3.4%)<br>18,887 (27.4%)<br>22,031 (32.0%)<br>213 (1.47) | 5,280 (20.8%)<br>867 (3.4%)<br>865 (3.4%)<br>6,996 (27.6%)<br>7,446 (29.4%)<br>2.18 (1.43) | -0.3% (-0.9%, 0.2%)<br>0.2% (-0.1%, 0.5%)<br>-0.0% (-0.3%, 0.2%)<br>-0.2% (-0.8%, 0.5%)<br>2.6% (1.9%, 3.3%)<br>-0.05 (-0.07, -0.03) | 5,355 (21.1%)<br>840 (3.3%)<br>854 (3.4%)<br>6,963 (27.5%)<br>7,498 (29.6%) | 3,296 (13.0%)<br>5,280 (20.8%)<br>867 (3.4%)<br>865 (3.4%)<br>6,993 (27.6%)<br>7,442 (29.4%) | 0.3% (-0.4%, 1.0%)<br>-0.1% (-0.4%, 0.2%)<br>-0.0% (-0.4%, 0.3%)<br>-0.1% (-0.9%, 0.7%)<br>0.2% (-0.6%, 1.0%)<br>-0.02 (-0.04, 0.01) |
| Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbA1C testsmean (sd)median [IQR]min, max Lipid panels | 14,120 (20.5%)<br>2,496 (3.6%)<br>2,335 (3.4%)<br>18,887 (27.4%)<br>22,031 (32.0%)<br>213 (1.47)<br>2.00 [1.00, 3.00]<br>0.00, 151.00 | 5,280 (20.8%)<br>867 (3.4%)<br>865 (3.4%)<br>6,996 (27.6%)<br>7,446 (29.4%)<br>218 (1.43)<br>2.00 [1.00, 3.00]<br>0.00, 66.00 | -0.3% (-0.9%, 0.2%)<br>0.2% (-0.13%, 0.5%)<br>-0.0% (-0.3%, 0.2%)<br>-0.2% (-0.8%, 0.5%)<br>2.6% (1.9%, 3.3%)<br>-0.05 (-0.07, -0.03)<br>-(-,-) | 5,355 (21.1%)<br>840 (3.3%)<br>854 (3.4%)<br>6,963 (27.5%)<br>7,498 (29.6%)<br>2.17 (1.36)<br>2.00 [1.00, 3.00]<br>0.00, 35.00 | 3.296 (13.0%) 5.280 (20.8%) 867 (3.4%) 865 (3.4%) 6.993 (27.6%) 7.442 (29.4%) 218 (1.41) 2.00 (1.00, 3.00) 0.00, 66.00 | 0.3% (-0.4%, 1.0%) -0.1% (-0.4%, 0.2%) -0.0% (-0.4%, 0.3%) -0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 1.0%) -0.02 (-0.04, 0.01) -(·, ·) -(·, ·) |
| Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbAIC testsmean (sd)median [IQR]min, max Lipid panelsmean (sd) | 14,120 (20.5%)<br>2,496 (3.6%)<br>2,335 (3.4%)<br>18,887 (27.4%)<br>22,031 (32.0%)<br>213 (1.47)<br>200 [1.00, 3.00]<br>0.00, 151.00 | 5,280 (20.8%)<br>867 (3.4%)<br>865 (3.4%)<br>6,996 (27.6%)<br>7,446 (29.4%)<br>218 (1.43)<br>200 [1.00, 3.00]<br>0.00, 66.00 | -0.3% (-0.9%, 0.2%) 0.2% (-0.1%, 0.5%) 0.2% (-0.3%, 0.2%) -0.2% (-0.8%, 0.5%) 2.6% (1.9%, 3.3%) -0.05 (-0.07, -0.03) -(, -) -(, -) -(, -) | 5,355 (21.1%)<br>840 (3.3%)<br>854 (3.4%)<br>6,963 (27.5%)<br>7,498 (29.6%)<br>2.17 (1.36)<br>2.00 (1.00, 3.00)<br>0.00, 35.00 | 3,296 (13.0%) 5,280 (20.8%) 867 (3.4%) 865 (3.4%) 6,993 (27.6%) 7,442 (29.4%) 218 (1.41) 200 [1.00, 3.00] 0.00, 66.00 | 0.3% (-0.4%, 1.0%) -0.1% (-0.4%, 0.2%) -0.0% (-0.4%, 0.3%) -0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 1.0%) -0.02 (-0.04, 0.01) -(-, -) -(-, -) -(-, -) |
| Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbA1C testsmean (sd)median [IQR]min, max Lipid panelsmean (sd)median [IQR]mening(sd)median [IQR] | 14,120 (20.5%)<br>2,496 (3.6%)<br>2,335 (3.4%)<br>18,887 (27.4%)<br>22,031 (32.0%)<br>213 (1.47)<br>200 (1.00, 3.00)<br>0.00,151.00<br>1.54 (1.27)<br>1.00 (1.00, 2.00) | 5,280 (20.8%)<br>867 (3.4%)<br>865 (3.4%)<br>6,996 (27.6%)<br>7,446 (29.4%)<br>218 (1.43)<br>2.00 [1.00, 3.00]<br>0.00, 66.00 | -0.3% (-0.9%, 0.2%) 0.2% (-0.1%, 0.5%) 0.2% (-0.3%, 0.2%) 0.2% (-0.8%, 0.5%) 2.6% (1.9%, 3.3%) -0.05 (-0.07, -0.03) -(-, -) -(-, -) -0.05 (-0.07, -0.03) -(-, -) | 5,355 (21.1%)<br>840 (3.3%)<br>854 (3.4%)<br>6,963 (27.5%)<br>7,498 (29.6%)<br>217 (1.36)<br>2.00 [1.00, 3.00]<br>0.00, 35.00<br>1.57 (1.15)<br>1.00 [1.00, 2.00] | 3,296 (13.0%) 5,280 (20.8%) 867 (3.4%) 865 (3.4%) 6,993 (27.6%) 7,442 (29.4%) 218 (1.41) 2.00 [1.00, 3.00] 0.00, 66.00 158 (1.17) 1.00 [1.00, 2.00] | 0.3% (-0.4%, 1.0%) -0.1% (-0.4%, 0.2%) -0.0% (-0.4%, 0.3%) -0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 1.0%) -0.02 (-0.04, 0.01) -(-, -) -(-, -) -0.01 (-0.03, 0.01) -(-, -) |
| Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbA1C testsmean (sd)median [IQR]min, max Lipid panelsmean (sd)median [IQR]median [IQR]median [IQR] | 14,120 (20.5%)<br>2,496 (3.6%)<br>2,335 (3.4%)<br>18,887 (27.4%)<br>22,031 (32.0%)<br>213 (1.47)<br>200 [1.00, 3.00]<br>0.00, 151.00 | 5,280 (20.8%)<br>867 (3.4%)<br>865 (3.4%)<br>6,996 (27.6%)<br>7,446 (29.4%)<br>218 (1.43)<br>200 [1.00, 3.00]<br>0.00, 66.00 | -0.3% (-0.9%, 0.2%) 0.2% (-0.1%, 0.5%) 0.2% (-0.3%, 0.2%) -0.2% (-0.8%, 0.5%) 2.6% (1.9%, 3.3%) -0.05 (-0.07, -0.03) -(, -) -(, -) -(, -) | 5,355 (21.1%)<br>840 (3.3%)<br>854 (3.4%)<br>6,963 (27.5%)<br>7,498 (29.6%)<br>2.17 (1.36)<br>2.00 (1.00, 3.00)<br>0.00, 35.00 | 3,296 (13.0%) 5,280 (20.8%) 867 (3.4%) 865 (3.4%) 6,993 (27.6%) 7,442 (29.4%) 218 (1.41) 200 [1.00, 3.00] 0.00, 66.00 | 0.3% (-0.4%, 1.0%) -0.1% (-0.4%, 0.2%) -0.0% (-0.4%, 0.3%) -0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 1.0%) -0.02 (-0.04, 0.01) -(-, -) -(-, -) -(-, -) |
| Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbA1C testsmean (sd)median [IQR]min, max Lipid panelsmean (sd)median [IQR]min, max Creatinine tests | 14,120 (20.5%) 2,496 (3.6%) 2,335 (3.4%) 18,887 (27.4%) 22,031 (32.0%) 213 (1.47) 2.00 (1.00, 3.00) 0.00, 151.00 1.54 (1.27) 1.00 (1.00, 2.00) 0.00, 149.00 | 5,280 (20.8%)<br>867 (3.4%)<br>865 (3.4%)<br>6,996 (27.6%)<br>7,446 (29.4%)<br>218 (1.43)<br>200 [1.00, 3.00]<br>0.00, 66.00<br>159 (1.18)<br>100 [1.00, 2.00]<br>0.00, 3.000 | -0.3% (-0.9%, 0.2%) 0.2% (-0.1%, 0.5%) -0.0% (-0.3%, 0.2%) -0.0% (-0.3%, 0.5%) 2.6% (1.9%, 3.3%) -0.05 (-0.07, -0.03) -(-,-) -0.05 (-0.07, -0.03) -(-,-) -(-,-) | 5,355 (21.1%) 840 (3.3%) 854 (3.4%) 6,963 (27.5%) 7,498 (29.6%) 2.17 (1.36) 2.00 (1.00, 3.00) 0.00, 35.00 1.57 (1.15) 1.00 [1.00, 2.00] 0.00, 34.00 | 3,296 (13.0%) 5,280 (20.8%) 867 (3.4%) 865 (3.4%) 6,993 (27.6%) 7,442 (29.4%) 218 (1.41) 200 (1.00, 3.00) 0.00, 66.00 1.58 (1.17) 1.00 (1.00, 2.00) 0.00, 29.00 | 0.3% (-0.4%, 1.0%) -0.1% (-0.4%, 0.2%) -0.0% (-0.4%, 0.3%) -0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 1.0%) -0.02 (-0.04, 0.01) -(-,-) -(-,-) -(-,-) -(-,-) -(-,-) |
| Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbAIC testsmean (sd)median [IQR]min, max Lipid panelsmean (sd)median [IQR]min max Creatinine testsmean (sd) | 14,120 (20.5%) 2,496 (3.6%) 18,887 (27.4%) 22,031 (32.0%) 213 (1.47) 200 (1.00, 3.00) 0.00, 151.00 1.54 (1.27) 1.00 (1.00, 2.00) 0.00, 149.00 0.04 (0.40) | 5,280 (20.8%) 867 (3.4%) 865 (3.4%) 6,996 (27.6%) 7,446 (29.4%) 218 (1.43) 200 [1.00, 3.00] 0.00, 66.00 159 (1.18) 1.00 [1.00, 2.00] 0.00, 30.00 0.03 (0.24) | -0.3% (-0.9%, 0.2%) 0.2% (-0.1%, 0.5%) 0.2% (-0.3%, 0.2%) 0.2% (-0.3%, 0.5%) 2.6% (1.9%, 3.3%) -0.05 (-0.07, -0.03) -(-, -) | 5,355 (21.1%) 840 (3.3%) 854 (3.4%) 6,963 (27.5%) 7,498 (29.6%) 217 (1.36) 2.00 [1.00, 3.00] 0.00, 35.00 1.57 (1.15) 1.00 [1.00, 2.00] 0.00, 34.00 0.03 (0.23) | 3,296 (13.0%) 5,280 (20.8%) 867 (3.4%) 865 (3.4%) 6,993 (27.6%) 7,442 (29.4%) 218 (1.41) 200 [1.00, 3.00] 0.00, 56.00 1.58 (1.17) 1.00 [1.00, 2.00] 0.00, 29.00 | 0.3% (-0.4%, 1.0%) -0.1% (-0.4%, 0.2%) -0.0% (-0.4%, 0.3%) -0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 1.0%) -0.02 (-0.04, 0.01) -(-, -) -(-, -) -0.01 (-0.03, 0.01) -(-, -) -(-, -) -(-, -) -0.00 (-0.00, 0.00) |
| Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbA1C testsmean (sd)median [IQR]min, max Lipid panelsmean (sd)median [IQR]min, max Cipatinine testsmean (sd)median [IQR]min, max Creatinine testsmean (sd)median [IQR]min, max | 14,120 (20.5%) 2,496 (3.6%) 2,335 (3.4%) 18,887 (27.4%) 22,031 (32.0%) 213 (1.47) 200 [1.00, 3.00] 0.00, 151.00 1.54 (1.27) 1.00 [1.00, 2.00] 0.00, 149.00 0.04 (0.40) 0.00 [0.00, 0.00] | 5,280 (20.8%) 867 (3.4%) 865 (3.4%) 865 (3.4%) 6,996 (27.6%) 7,446 (29.4%) 218 (1.43) 200 [1.00, 3.00] 0.00, 66.00 1.59 (1.18) 1.00 [1.00, 2.00] 0.00, 30.00 0.03 (0.24) 0.00 [0.00, 0.00] | -0.3% (-0.9%, 0.2%) 0.2% (-0.1%, 0.5%) 0.2% (-0.3%, 0.2%) -0.2% (-0.8%, 0.5%) 2.6% (1.9%, 3.3%) -0.05 (-0.07, -0.03) -(-, -) | 5,355 (21.1%) 840 (3.3%) 854 (3.4%) 6,963 (27.5%) 7,498 (29.6%) 217 (1.36) 2.00 (1.00, 3.00) 0.00, 35.00 1.57 (1.15) 1.00 (1.00, 2.00) 0.00, 34.00 0.03 (0.23) 0.00 (0.00, 0.00) | 3,296 (13.0%) 5,280 (20.8%) 867 (3.4%) 865 (3.4%) 6,993 (27.6%) 7,442 (29.4%) 218 (1.41) 200 [1.00, 3.00] 0.00, 66.00 158 (1.17) 1.00 [1.00, 2.00] 0.00, 29.00 0.03 (0.24) 0.00 [0.00, 0.00] | 0.3% (-0.4%, 1.0%) -0.1% (-0.4%, 0.2%) -0.0% (-0.4%, 0.3%) -0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 1.0%) -0.02 (-0.04, 0.01) -(-, -) -(-, -) -0.01 (-0.03, 0.01) -(-, -) -0.00 (-0.00, 0.00) -(-, -) |
| Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbA1C testsmean (sd)median [IQR]min, max Lipid panelsmean (sd)median [IQR]min, max Cipid panelsmean (sd)median (IQR)min, max | 14,120 (20.5%) 2,496 (3.6%) 18,887 (27.4%) 22,031 (32.0%) 213 (1.47) 200 (1.00, 3.00) 0.00, 151.00 1.54 (1.27) 1.00 (1.00, 2.00) 0.00, 149.00 0.04 (0.40) | 5,280 (20.8%) 867 (3.4%) 865 (3.4%) 6,996 (27.6%) 7,446 (29.4%) 218 (1.43) 200 [1.00, 3.00] 0.00, 66.00 159 (1.18) 1.00 [1.00, 2.00] 0.00, 30.00 0.03 (0.24) | -0.3% (-0.9%, 0.2%) 0.2% (-0.1%, 0.5%) 0.2% (-0.3%, 0.2%) 0.2% (-0.3%, 0.5%) 2.6% (1.9%, 3.3%) -0.05 (-0.07, -0.03) -(-, -) | 5,355 (21.1%) 840 (3.3%) 854 (3.4%) 6,963 (27.5%) 7,498 (29.6%) 217 (1.36) 2.00 [1.00, 3.00] 0.00, 35.00 1.57 (1.15) 1.00 [1.00, 2.00] 0.00, 34.00 0.03 (0.23) | 3,296 (13.0%) 5,280 (20.8%) 867 (3.4%) 865 (3.4%) 6,993 (27.6%) 7,442 (29.4%) 218 (1.41) 200 [1.00, 3.00] 0.00, 56.00 1.58 (1.17) 1.00 [1.00, 2.00] 0.00, 29.00 | 0.3% (-0.4%, 1.0%) -0.1% (-0.4%, 0.2%) -0.0% (-0.4%, 0.3%) -0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 1.0%) -0.02 (-0.04, 0.01) -(-, -) -(-, -) -0.01 (-0.03, 0.01) -(-, -) -(-, -) -(-, -) -0.00 (-0.00, 0.00) |
| Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbAIC testsmean (sd)median [IQR]min, max Lipid panelsmean (sd)median [IQR]min, max Creatinine testsmean (sd)median [IQR]min, max Creatinine testsmean (sd)median [IQR]min, max Creatinine testsmean (sd)median [IQR]min, max Natiuretic peptide tests | 14,120 (20.5%) 2,496 (3.6%) 2,335 (3.4%) 18,887 (27.4%) 22,031 (32.0%) 213 (1.47) 2.00 [1.00, 3.00] 0.00, 151.00 1.54 (1.27) 1.00 [1.00, 2.00] 0.00, 149.00 0.04 (0.40) 0.00 [0.00, 0.00] 0.00, 43.00 | 5,280 (20.8%) 867 (3.4%) 867 (3.4%) 6,996 (27.6%) 7,446 (29.4%) 218 (1.43) 200 [1.00, 3.00] 0.00, 66.00 1.59 (1.18) 1.00 [1.00, 2.00] 0.00, 30.00 0.03 (0.24) 0.00 [0.00, 0.00] 0.00, 10.00 | -0.3% (-0.9%, 0.2%) 0.2% (-0.1%, 0.5%) 0.2% (-0.3%, 0.2%) 0.2% (-0.3%, 0.5%) 2.6% (1.9%, 3.3%) -0.05 (-0.07, -0.03) -(-, -) | 5,355 (21.1%) 840 (3.3%) 854 (3.4%) 6,963 (27.5%) 7,498 (29.6%) 2.17 (1.36) 2.00 [1.00, 3.00] 0.00, 35.00 1.57 (1.15) 1.00 [1.00, 2.00] 0.00, 34.00 0.03 (0.23) 0.00 [0.00, 0.00] 0.00, 10.00 | 3,296 (13.0%) 5,280 (20.8%) 867 (3.4%) 865 (3.4%) 6,993 (27.6%) 7,442 (29.4%) 218 (1.41) 200 [1.00, 3.00] 0.00, 66.00 1.58 (1.17) 1.00 [1.00, 2.00] 0.00, 29.00 0.03 (0.24) 0.00 [0.00, 0.00] 0.00, 10.00 | 0.3% (-0.4%, 1.0%) -0.1% (-0.4%, 0.2%) -0.0% (-0.4%, 0.3%) -0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 1.0%) -0.02 (-0.04, 0.01) -(-, -) |
| Fecal occult blood test; n (%) Bone mineral densify tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbA1C testsmean (sd)median [IQR]min, max Lipid panelsmean (sd)median [IQR]min, max Creatinine testsmean (sd)median [IQR]min, max Creatinine testsmean (sd)median [IQR]min, max Arriver (sd)median [IQR]min, max Arriver (sd)median [IQR]min, max Arriver (sd)median [IQR]min, max Arriver (sd)median [IQR]min, max Arriver (sd)median (sd) | 14,120 (20.5%) 2,496 (3.6%) 2,335 (3.4%) 18,887 (27.4%) 22,031 (32.0%) 213 (1.47) 200 (1.00, 3.00) 0.00, 151.00 1.54 (1.27) 1.00 [1.00, 2.00] 0.00, 149.00 0.04 (0.40) 0.00 [0.00, 0.00] 0.00, 43.00 0.11 (0.77) | 5,280 (20.8%) 867 (3.4%) 865 (3.4%) 6,996 (27.6%) 7,446 (29.4%) 218 (1.43) 2.00 (1.00, 3.00) 0.00, 66.00 1.59 (1.18) 1.00 (1.00, 2.00) 0.00, 30.00 0.03 (0.24) 0.00 (0.00, 0.00) 0.00, 10.00 0.10 (0.60) | -0.3% (-0.9%, 0.2%) 0.2% (-0.1%, 0.5%) 0.2% (-0.3%, 0.2%) 0.2% (-0.8%, 0.5%) 2.6% (1.9%, 3.3%) -0.05 (-0.07, -0.03) -(-, -) | 5,355 (21.1%) 840 (3.3%) 854 (3.4%) 6,963 (27.5%) 7,498 (29.6%) 217 (1.36) 2.00 [1.00, 3.00] 0.00, 35.00 1.57 (1.15) 1.00 [1.00, 2.00] 0.00, 34.00 0.03 (0.23) 0.00 [0.00, 0.00] 0.00, 10.00 0.10 (0.65) | 3,296 (13.0%) 5,280 (20.8%) 867 (3.4%) 865 (3.4%) 6,993 (27.6%) 7,442 (29.4%) 218 (1.41) 200 [1.00, 3.00] 0.00, 66.00 1.58 (1.17) 1.00 [1.00, 2.00] 0.00, 29.00 0.03 (0.24) 0.00 [0.00, 0.00] 0.00, 10.00 0.10 (0.60) | 0.3% (-0.4%, 1.0%) -0.1% (-0.4%, 0.2%) -0.0% (-0.4%, 0.3%) -0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 1.0%) -(-, -) |
| Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbA1C testsmean (sd)median [IQR]min, max Lipid panelsmean (sd)median [IQR]min, max Creatinine testsmean (sd)median [IQR]min, max Variuretic peptide testsmean (sd)median [IQR]min, max | 14,120 (20.5%) 2,496 (3.6%) 2,335 (3.4%) 18,887 (27.4%) 22,031 (32.0%) 213 (1.47) 200 (1.00, 3.00) 0.00, 151.00 1.54 (1.27) 1.00 (1.00, 2.00) 0.00, 149.00 0.04 (0.40) 0.00 (0.00, 0.00) 0.00, 43.00 0.11 (0.77) 0.00 [0.00, 0.00] | 5,280 (20.8%) 867 (3.4%) 865 (3.4%) 865 (3.4%) 6,996 (27.6%) 7,446 (29.4%) 218 (1.43) 2.00 [1.00, 3.00] 0.00, 66.00 1.59 (1.18) 1.00 [1.00, 2.00] 0.00, 3.0.00 0.03 (0.24) 0.00 [0.00, 0.00] 0.00, 10.00 0.10 (0.60) 0.00 [0.00, 0.00] | -0.3% (-0.9%, 0.2%) 0.2% (-0.1%, 0.5%) 0.2% (-0.3%, 0.2%) -0.2% (-0.8%, 0.5%) 2.6% (1.9%, 3.3%) -0.05 (-0.07, -0.03) -(-, -) | 5,355 (21.1%) 840 (3.3%) 854 (3.4%) 6,963 (27.5%) 7,498 (29.6%) 217 (1.36) 200 (1.00, 3.00) 0.00, 35.00 1.57 (1.15) 1.00 (1.00, 2.00) 0.00, 34.00 0.03 (0.23) 0.00 (0.00, 0.00) 0.00 (0.00) 0.01 (0.65) 0.00 (0.00, 0.00) | 3,296 (13.0%) 5,280 (20.8%) 867 (3.4%) 865 (3.4%) 6,993 (27.6%) 7,442 (29.4%) 218 (1.41) 200 [1.00, 3.00] 0.00, 66.00 1.58 (1.17) 1.00 [1.00, 2.00] 0.00, 29.00 0.03 (0.24) 0.00 [0.00, 0.00] 0.00, 10.00 0.10 (0.60) 0.10 (0.60) 0.00 [0.00, 0.00] | 0.3% (-0.4%, 1.0%) -0.1% (-0.4%, 0.2%) -0.0% (-0.4%, 0.3%) -0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 1.0%) -0.02 (-0.04, 0.01) -(-, -) -(-, -) -(-, -) -0.01 (-0.03, 0.01) -(-, -) |
| Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbA1C testsmean (sd)median [IQR]min, max Lipid panelsmean (sd)median [IQR]min, max Creatinine testsmean (sd)mean (sd)min, max Variante (sd)mean (sd) | 14,120 (20.5%) 2,496 (3.6%) 2,335 (3.4%) 18,887 (27.4%) 22,031 (32.0%) 213 (1.47) 200 (1.00, 3.00) 0.00, 151.00 1.54 (1.27) 1.00 [1.00, 2.00] 0.00, 149.00 0.04 (0.40) 0.00 [0.00, 0.00] 0.00, 43.00 0.11 (0.77) | 5,280 (20.8%) 867 (3.4%) 865 (3.4%) 6,996 (27.6%) 7,446 (29.4%) 218 (1.43) 2.00 (1.00, 3.00) 0.00, 66.00 1.59 (1.18) 1.00 (1.00, 2.00) 0.00, 30.00 0.03 (0.24) 0.00 (0.00, 0.00) 0.00, 10.00 0.10 (0.60) | -0.3% (-0.9%, 0.2%) 0.2% (-0.1%, 0.5%) 0.2% (-0.3%, 0.2%) 0.2% (-0.8%, 0.5%) 2.6% (1.9%, 3.3%) -0.05 (-0.07, -0.03) -(-, -) | 5,355 (21.1%) 840 (3.3%) 854 (3.4%) 6,963 (27.5%) 7,498 (29.6%) 217 (1.36) 2.00 [1.00, 3.00] 0.00, 35.00 1.57 (1.15) 1.00 [1.00, 2.00] 0.00, 34.00 0.03 (0.23) 0.00 [0.00, 0.00] 0.00, 10.00 0.10 (0.65) | 3,296 (13.0%) 5,280 (20.8%) 867 (3.4%) 865 (3.4%) 6,993 (27.6%) 7,442 (29.4%) 218 (1.41) 200 [1.00, 3.00] 0.00, 66.00 1.58 (1.17) 1.00 [1.00, 2.00] 0.00, 29.00 0.03 (0.24) 0.00 [0.00, 0.00] 0.00, 10.00 0.10 (0.60) | 0.3% (-0.4%, 1.0%) -0.1% (-0.4%, 0.2%) -0.0% (-0.4%, 0.3%) -0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 1.0%) -(-, -) |
| Fecal occult blood test n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbA1C testsmean (sd)median [IQR]min, max Lipid panelsmean (sd)median [IQR]min, max Creatinine testsmean (sd)median [IQR]min, max Mammograms Mammogra | 14,120 (20.5%) 2,496 (3.6%) 2,335 (3.4%) 18,887 (27.4%) 22,031 (32.0%) 213 (1.47) 2.00 [1.00, 3.00] 0.00, 151.00 1.54 (1.27) 1.00 [1.00, 2.00] 0.00, 149.00 0.04 (0.40) 0.00 [0.00, 0.00] 0.00, 43.00 0.11 (0.77) 0.00 [0.00, 0.00] 0.00, 62.00 | 5,280 (20.8%) 867 (3.4%) 865 (3.4%) 6,996 (27.6%) 7,446 (29.4%) 218 (1.43) 200 [1.00, 3.00] 0.00, 66.00 1.59 (1.18) 1.00 [1.00, 2.00] 0.00, 30.00 0.03 (0.24) 0.00 (0.00, 0.00] 0.00, 10.00 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 0.00, 28.00 | -0.3% (-0.9%, 0.2%) 0.2% (-0.1%, 0.5%) 0.2% (-0.3%, 0.2%) 0.2% (-0.3%, 0.5%) 2.6% (1.9%, 3.3%) -0.05 (-0.07, -0.03) -(-, -) | 5,355 (21.1%) 840 (3.3%) 840 (3.3%) 6,963 (27.5%) 7,498 (29.6%) 217 (1.36) 2.00 [1.00, 3.00] 0.00, 35.00 1.57 (1.15) 1.00 [1.00, 2.00] 0.00, 34.00 0.03 (0.23) 0.00 [0.00, 0.00] 0.00, 10.00 0.10 (0.65) 0.00 [0.00, 0.00] 0.00, 27.00 | 3,296 (13.0%) 5,280 (20.8%) 867 (3.4%) 865 (3.4%) 6,993 (27.6%) 7,442 (29.4%) 218 (1.41) 2.00 (1.00, 3.00) 0.00, 66.00 1.58 (1.17) 1.00 (1.00, 2.00) 0.00, 29.00 0.03 (0.24) 0.00 (0.00, 0.00) 0.00 (0.00, 0.00) 0.00 (0.00, 0.00) 0.00 (0.00, 0.00) 0.00 (0.00, 0.00) 0.00, 28.00 | 0.3% (-0.4%, 1.0%) -0.1% (-0.4%, 0.2%) -0.0% (-0.4%, 0.3%) -0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 1.0%) -0.02 (-0.04, 0.01) -(-, -) |
| Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbA1C testsmean (sd)median [IQR]min, max Lipid panelsmean (sd)median [IQR]min, max Creatinine testsmean (sd)median [IQR]min, max Notatinine testsmean (sd)median [IQR]min, max Matriuretic peptide testsmean (sd)median [IQR]min, max Undian [IQR]min, max Undian [IQR]min, max Undian [IQR]min, max University sets setsmean (sd)median [IQR]min, max University setsmedian [IQR]min, max University setsmedian [IQR]min, max University setsmean (sd)median [IQR]min, max University setsmean (sd) | 14,120 (20.5%) 2,496 (3.6%) 2,335 (3.4%) 18,887 (27.4%) 22,031 (32.0%) 213 (1.47) 2.00 [1.00, 3.00] 0.00, 151.00 1.54 (1.27) 1.00 [1.00, 2.00] 0.00, 149.00 0.04 (0.40) 0.00 [0.00, 0.00] 0.00, 43.00 0.11 (0.77) 0.00 [0.00, 0.00] 0.00, 62.00 0.90 (1.60) | 5,280 (20.8%) 867 (3.4%) 865 (3.4%) 865 (3.4%) 6,996 (27.6%) 7,446 (29.4%) 218 (1.43) 2.00 [1.00, 3.00] 0.00, 66.00 1.59 (1.18) 1.00 [1.00, 2.00] 0.00, 30.00 0.03 (0.24) 0.00 [0.00, 0.00] 0.00, 10.00 0.10 (0.60) 0.00 [0.00, 0.00] 0.00, 28.00 0.867 (3.4%) | -0.3% (-0.9%, 0.2%) 0.2% (-0.1%, 0.5%) -0.0% (-0.3%, 0.2%) -0.2% (-0.8%, 0.5%) 2.6% (1.9%, 3.3%) -0.05 (-0.07, -0.03) -(-, -) | 5,355 (21.1%) 840 (3.3%) 854 (3.4%) 6,963 (27.5%) 7,498 (29.6%) 217 (1.36) 2.00 [1.00, 3.00] 0.00, 35.00 1.57 (1.15) 1.00 [1.00, 2.00] 0.00, 34.00 0.03 (0.23) 0.00 [0.00, 0.00] 0.00, 10.00 0.10 (0.65) 0.00 [0.00, 0.00] 0.00, 27.00 0.89 (1.54) | 3,296 (13.0%) 5,280 (20.8%) 865 (3.4%) 865 (3.4%) 6,993 (27.6%) 7,442 (29.4%) 218 (1.41) 200 [1.00, 3.00] 0.00, 66.00 1.58 (1.17) 1.00 [1.00, 2.00] 0.00, 29.00 0.03 (0.24) 0.00 [0.00, 0.00] 0.00 [0.00, 0.00] 0.00 [0.00, 0.00] 0.00 [0.00, 0.00] 0.00, 28.00 | 0.3% (-0.4%, 1.0%) -0.1% (-0.4%, 0.2%) -0.0% (-0.4%, 0.3%) -0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 1.0%) -(-, -) |
| Fecal occult blood test; n (%) Bone mineral density tests; n (%) Mammograms; n (%) Telemedicine; n (%) HbA1C testsmean (sd)median [IQR]min, max Lipid panelsmean (sd)median [IQR]min, max Creatinine testsmean (sd)median [IQR]min, max Creatinine testsmean (sd)median [IQR]min, max Naturetic peptide testsmean (sd)median [IQR]min, max Natriuretic peptide testsmean (sd)median [IQR]min, max Urine testsmean (sd)median [IQR]min, max Urine tests | 14,120 (20.5%) 2,496 (3.6%) 2,335 (3.4%) 18,887 (27.4%) 22,031 (32.0%) 213 (1.47) 2.00 [1.00, 3.00] 0.00, 151.00 1.54 (1.27) 1.00 [1.00, 2.00] 0.00, 149.00 0.04 (0.40) 0.00 [0.00, 0.00] 0.00, 43.00 0.11 (0.77) 0.00 [0.00, 0.00] 0.00, 62.00 | 5,280 (20.8%) 867 (3.4%) 865 (3.4%) 6,996 (27.6%) 7,446 (29.4%) 218 (1.43) 200 [1.00, 3.00] 0.00, 66.00 1.59 (1.18) 1.00 [1.00, 2.00] 0.00, 30.00 0.03 (0.24) 0.00 (0.00, 0.00] 0.00, 10.00 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 0.00 (0.00, 0.00] 0.00, 28.00 | -0.3% (-0.9%, 0.2%) 0.2% (-0.1%, 0.5%) 0.2% (-0.3%, 0.2%) 0.2% (-0.3%, 0.5%) 2.6% (1.9%, 3.3%) -0.05 (-0.07, -0.03) -(-, -) | 5,355 (21.1%) 840 (3.3%) 840 (3.3%) 6,963 (27.5%) 7,498 (29.6%) 217 (1.36) 2.00 [1.00, 3.00] 0.00, 35.00 1.57 (1.15) 1.00 [1.00, 2.00] 0.00, 34.00 0.03 (0.23) 0.00 [0.00, 0.00] 0.00, 10.00 0.10 (0.65) 0.00 [0.00, 0.00] 0.00, 27.00 | 3,296 (13.0%) 5,280 (20.8%) 867 (3.4%) 865 (3.4%) 6,993 (27.6%) 7,442 (29.4%) 218 (1.41) 2.00 (1.00, 3.00) 0.00, 66.00 1.58 (1.17) 1.00 (1.00, 2.00) 0.00, 29.00 0.03 (0.24) 0.00 (0.00, 0.00) 0.00 (0.00, 0.00) 0.00 (0.00, 0.00) 0.00 (0.00, 0.00) 0.00 (0.00, 0.00) 0.00, 28.00 | 0.3% (-0.4%, 1.0%) -0.1% (-0.4%, 0.2%) -0.0% (-0.4%, 0.3%) -0.1% (-0.9%, 0.7%) 0.2% (-0.6%, 1.0%) -0.02 (-0.04, 0.01) -(-, -) |

| Combined comorbidity score | | | | | | |
|---|---|---|---|---|---|---|
| mean (sd) | 0.98 (1.67) | 0.92 (1.57) | 0.06 (0.04, 0.08) | 0.93 (1.61) | 0.92 (1.57) | 0.01 (-0.02, 0.03) |
| median [IQR] | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | - (-, -) | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | - (-, -) |
| min, max | -2.00, 17.00 | -2.00, 14.00 | - (-, -) | -2.00, 13.00 | -2.00, 14.00 | - (-, -) |
| Frailty Score | | | | | | |
| mean (sd) | 0.14 (0.04) | 0.14 (0.04) | 0.00 (0.00, 0.00) | 0.14 (0.04) | 0.14 (0.04) | -0.00 (-0.00, 0.00) |
| median [IQR] | 0.13 [0.12, 0.16] | 0.13 [0.12, 0.16] | - (-, -) | 0.13 [0.12, 0.16] | 0.13 [0.12, 0.16] | - (-, -) |
| min, max | 0.04, 0.56 | 0.04, 0.49 | - (-, -) | 0.04, 0.56 | 0.04, 0.49 | - (-, -) |
| Number of Hospitalizations | | | | | | |
| mean (sd) | 4.49 (26.85) | 3.77 (20.18) | 0.72 (0.40, 1.04) | 3.86 (20.72) | 3.76 (20.06) | 0.10 (-0.25, 0.46) |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) |
| min, max | 0.00, 3,896.00 | 0.00, 627.00 | - (-, -) | 0.00, 733.00 | 0.00, 627.00 | - (-, -) |
| Any hospitalization within prior 91 days; n (%) | 1,844 (2.7%) | 578 (2.3%) | 0.4% (0.2%, 0.6%) | 596 (2.4%) | 578 (2.3%) | 0.1% (-0.2%, 0.3%) |
| Any hospitalization within prior 92-365 days; n (%) | 4,068 (5.9%) | 1,299 (5.1%) | 0.8% (0.5%, 1.1%) | 1,293 (5.1%) | 1,298 (5.1%) | -0.0% (-0.4%, 0.4%) |
| Number of hospitalizations (0, 1, 2 or more) | | | | | | |
| < 1; n (%) | 63,460 (92.1%) | 23,628 (93.2%) | -1.1% (-1.5%, -0.7%) | 23,616 (93.2%) | 23,618 (93.2%) | -0.0% (-0.5%, 0.4%) |
| 1 - <2; n (%) | 444 (0.6%) | 138 (0.5%) | 0.1% (-0.0%, 0.2%) | 142 (0.6%) | 138 (0.5%) | 0.0% (-0.1%, 0.1%) |
| >= 2; n (%) | 5,028 (7.3%) | 1,591 (6.3%) | 1.0% (0.7%, 1.4%) | 1,588 (6.3%) | 1,590 (6.3%) | -0.0% (-0.4%, 0.4%) |
| Heart failure hospitalization; n (%) | 1,204 (1.7%) | 325 (1.3%) | 0.5% (0.3%, 0.6%) | 341 (1.3%) | 325 (1.3%) | 0.1% (-0.1%, 0.3%) |
| ED visit; n (%) | 19,883 (28.8%) | 6,921 (27.3%) | 1.6% (0.9%, 2.2%) | 7,010 (27.7%) | 6,918 (27.3%) | 0.4% (-0.4%, 1.1%) |
| Acute MI; n (%) | 593 (0.9%) | 182 (0.7%) | 0.1% (0.0%, 0.3%) | 182 (0.7%) | 182 (0.7%) | 0.0% (-0.1%, 0.1%) |
| Old MI; n (%) | 1,038 (1.5%) | 280 (1.1%) | 0.4% (0.2%, 0.6%) | 269 (1.1%) | 280 (1.1%) | -0.0% (-0.2%, 0.1%) |
| Heart failure; n (%) | 3,822 (5.5%) | 1,182 (4.7%) | 0.9% (0.6%, 1.2%) | 1,227 (4.8%) | 1,181 (4.7%) | 0.2% (-0.2%, 0.6%) |
| Acute heart failure; n (%) | 970 (1.4%) | 248 (1.0%) | 0.4% (0.3%, 0.6%) | 254 (1.0%) | 247 (1.0%) | 0.0% (-0.1%, 0.2%) |
| Microalbuminuria or proteinuria; n (%) | 2,327 (3.4%) | 825 (3.3%) | 0.1% (-0.1%, 0.4%) | 825 (3.3%) | 825 (3.3%) | 0.0% (-0.3%, 0.3%) |
| Ratio of brand to generic medications | | | | | | |
| mean (sd) | 1.02 (0.04) | 1.01 (0.04) | 0.00 (0.00, 0.00) | 1.01 (0.04) | 1.01 (0.04) | -0.00 (-0.00, 0.00) |
| median [IQR] | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | - (-, -) | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | - (-, -) |
| min, max | 0.80, 2.00 | 0.83, 1.43 | - (-, -) | 0.80, 1.50 | 0.83, 1.43 | - (-, -) |

Variable\_name

Gender Race

Region

Smoking / Tobacco use Underweight Normal weight, if BMI is 20.0-24.9

Overweight, if BMI is 25.0 to 29.9 Class 1 (low-risk) obesity, if BMI is 30.0 to 34.9 Class 2 (moderate-risk) obesity, if BMI is 35.0 to 39.9 Class 3 (high-risk) obesity if BMI is equal to or greater than 40

Unspecified obesity Diabetic retinopathy

Diabetic neuropathy Diabetic nephropathy

Diabetes with other opthalmic complications

Diabetes with peripheral circulatory disorders

Diabetic foot

Erectile dysfuntion

Hypoglycemia

Hyperglycemia/DKA/HONK

Skin infections

Stable angina

Unstable angina

Hypertension

Hypotension

Hyperlipidemia Atrial fibrillation Acute myocardial infarction Old myocardial infarction

Cardiac conduction disorder

Previous cardiac procedure (CABG, PTCA, Stent)

Ischemic stroke PVD diagnosis or surgery

Other cardiac dysrhythmia

Heart failure

Acute heart failure

Microalbuminuria/proteinuria

#### Algorithm sources

If region not available, from State, https://www2.census.gov/geo/pdfs/mapsdata/maps/reference/us\_regdiv.pdf

Investigator review of codes based on:

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015.

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002.

https://pubmed.ncbi.nlm.nih.gov/34953068/.

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9154288/.

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3721171/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/,

https://pubmed.ncbi.nlm.nih.gov/35043165/ Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/,

https://pubmed.ncbi.nlm.nih.gov/35043165/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/ Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/, ICD9 to ICD10 conversion

Investigator review of codes based on:

https://www.ncbi.nlm.nih.gov/books/NBK368403/table/sb203.t5/,

https://www.health.mil/Reference-Center/Publications/2016/03/01/Diabetes-Mellitus,

http://www.icd9data.com/2014/Volume1/240-279/249-259/250/default.htm,

https://www.icd10data.com/ICD10CM/Codes/E00-E89/E08-E13/E11-

Intps://www.icd10data.com/ICD10CM/Codes/N00-N99/N40-N53/N52-,

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4857901/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/,

https://pubmed.ncbi.nlm.nih.gov/35043165/

Investigator review of codes based on:

Hyperglycemia: https://pubmed.ncbi.nlm.nih.gov/34953068/.

https://pubmed.ncbi.nlm.nih.gov/35043165/

DKA: https://pubmed.ncbi.nlm.nih.gov/29773640/. https://pubmed.ncbi.nlm.nih.gov/38262528/

https://dam.assets.ohio.gov/image/upload/medicaid.ohio.gov/Providers/PaymentInnovatio n/DEF/DKA.pdf

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/ . ICD9 to ICD10 conversion

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/19337843/,

https://pmc.ncbi.nlm.nih.gov/articles/PMC9172873/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/19337843/, https://pmc.ncbi.nlm.nih.gov/articles/PMC9172873/ Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/,

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8929186/

Investigator review of codes based on: https://pmc.ncbi.nlm.nih.gov/articles/PMC8064679/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/,

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002,

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/31933524/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/24682186/ Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/24682186/ Investigator review of codes based on:

https://stacks.cdc.gov/view/cdc/31381/cdc\_31381\_DS8.pdf,

https://www.health.ny.gov/health\_care/medicaid/redesign/dsrip/vbp\_library/docs/arrblk.p

df, https://www.cdc.gov/dhdsp/maps/atlas/data-sources.html,

https://www.cms.gov/medicare/coding/icd10/downloads/icd10clinicalconceptscardiology

1.pdf, ICD9 to ICD10 conversion

Modified codes based on eligibility criteria, here we implement any care setting, any diagnosis position

Modified codes based on eligibility criteria, here we implement any care setting, any diagnosis position

Investigator review of codes, https://www.icd10data.com/

Investigator review of codes based on:

 $https://stacks.cdc.gov/view/cdc/31381/cdc\_31381\_DS8.pdf,\\$ 

https://www.health.ny.gov/health\_care/medicaid/redesign/dsrip/vbp\_library/docs/arrblk.pdf, https://www.cdc.gov/dhdsp/maps/atlas/data-sources.html,

https://www.cms.gov/medicare/coding/icd10/downloads/icd10clinicalconceptscardiology

1.pdf, ICD9 to ICD10 conversion

Modified codes based on inclusion criteria, here we implement any care setting, any

diagnosis position Modified codes based on inclusion criteria, here we implement any care setting, any diagnosis position

Modified codes based on inclusion criteria, here we implement any care setting, any

diagnosis position

Cardiomyopathy Valve disorders Valve replacement TIA Edema Venous thromboembolism/ pulmonary embolsim Pulmonary hypertension Implantable cardioverter defibrillator Hyperkalemia Coronary atherosclerosis Cerebrovascular procedure Insertion of pacemakers / removal of cardiac lead CKD stage 1-2 CKD stage 3-4

Hypertensive nephropathy

Unspecified CKD Acute kidney injury

Urinary tract infections Genital infections

Urolithiasis (kidney or urinary stones)

COPD

Asthma

Obstructive sleep apnea

Serious bacterial infections

Pneumonia

Liver disease

MASH/MASLD

Fractures / Falls

Osteoporosis Osteoarthritis Depression

Dementia

Delirium or psychosis

Anxiety

Sleep disorder

Anemia Influenza

COVID-19

Investigator review of codes based on:

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder mpl2p wn015

Investigator review of codes based on:

https://stacks.cdc.gov/view/cdc/31381/cdc\_31381\_DS8.pdf,

https://pubmed.ncbi.nlm.nih.gov/38440888/

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8751938/,

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015,

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=cder\_mpl2p\_wp009 Modified codes based on eligibility criteria, here we implement any care setting, any diagnosis position

Modified codes based on eligibility criteria, here we implement any care setting, any

diagnosis position

Investigator review of codes based on: https://www.cms.gov/medicare-coveragedatabase/view/article.aspx?articleid=52993&ver=45&

Investigator review of codes based on:

https://www.sciencedirect.com/science/article/pii/S2666572723000251

Investigator review of codes

Modified codes based on eligibility criteria, here we implement any care setting, any diagnosis position

https://pmc.ncbi.nlm.nih.gov/articles/PMC4399109/

Investigator review of codes based on:

https://pmc.ncbi.nlm.nih.gov/articles/PMC10251803/

Investigator review of codes, https://www.icd10data.com/

Modified codes based on eligibility criteria, here we implement any care setting, any diagnosis position

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/

Investigator review of codes based on:

https://pmc.ncbi.nlm.nih.gov/articles/PMC2978782/ Investigator review of codes based on:

https://pmc.ncbi.nlm.nih.gov/articles/PMC5888226/ Investigator review of codes based on:

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8929186/

Investigator review of codes based on:

https://nccd.cdc.gov/ckd/Methods.aspx?Qnum=Q637,

https://www.kidneymedicinejournal.org/cms/10.1016/j.xkme.2022.100414/attachment/5e/second-complex and the complex and the co29ab67-7a7d-4621-9af3-81bd071bbc67/mmc1.pdf,

https://www.icd10data.com/ICD10CM/Codes/I00-I99

Investigator reviewed code based on:

https://pmc.ncbi.nlm.nih.gov/articles/PMC7558992/#app1-antibiotics-09-00536

Investigator reviewed codes based on: https://pubmed.ncbi.nlm.nih.gov/30207042/

Investigator review of codes based on:

https://pmc.ncbi.nlm.nih.gov/articles/PMC7793999/

Investigator review of codes based on:

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10203971/

Investigator review of codes based on:

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10203971/, modified CCW algorithm (any

care setting, any diagnosis position)
Investigator review of codes based on:

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8636332/,

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7927325/

https://pubmed.ncbi.nlm.nih.gov/29921683/, https://pubmed.ncbi.nlm.nih.gov/17346615/,

https://pubmed.ncbi.nlm.nih.gov/23335588/

Investigator review of codes based on:

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10203971/

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002\_ https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015, Modified algorightm from\_

https://pubmed.ncbi.nlm.nih.gov/34256144/\_Modified.CCW\_algorithm Investigator review of codes: https://pubmed.ncbi.nlm.nih.gov/32300995/\_

https://pubmed.ncbi.nlm.nih.gov/39316292/

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015,

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

 $packages/browse? at = cder\_mpl2p\_wp009,$ 

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=cder\_mpl2p\_wp010

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8202643/,

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002, CCW Algorithms

Modified CCW algorithm

https://pubmed.ncbi.nlm.nih.gov/35043165/, CCW Algorithms

https://pubmed.ncbi.nlm.nih.gov/35043165/,

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015

https://pubmed.ncbi.nlm.nih.gov/28485014/, https://pubmed.ncbi.nlm.nih.gov/35043165/ ://pubmed.ncbi.nlm.nih.gov/35043165

Investigator review of codes based on https://www.verywellhealth.com/sleeping-disorders-list-anddiagnostic-codes-3014779

Modified codes based on eligibility criteria, here we implement any care setting, any diagnosis position

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/38556924/ https://pubmed.ncbi.nlm.nih.gov/34913208/,

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8427377/

Hyperthyroidism and other thyroid gland disorders

Hypothyroidism

Nephrotic syndrome Urinary incontinence

Biliary disease

Pancreatitis

Bowel obstruction Gastroparesis Number of antidiabetic drugs on CED

Concomitant use or initiation of metformin Concomitant use or initiation of insulin

Concomitant use or initiation of sulfonylureas

Concomitant use or initiation of DPP4i

Concomitant use or initiation of SGLT2i

Concomitant use or initiation of other glucose-lowering drugs

Past use of metformin

Past use of insulin

Past use of sulfonylureas

Past use of DPP4i

Past use of SGLT2i

Past use of other glucose-lowering drugs

ACEi / ARB

ARNI

Thiazides

Beta-Blockers

Calcium channel blockers

Digoxin / Digitoxin

Loop diuretics

Other diuretics Intravenous diuretics

Nitrates

Anti-arrhythmics

Statins

PCSK9 inhibitors and other lipid-lowering drugs

Antiplatelet agents

Oral anticoagulants

COPD/Asthma medication

NSAIDs

Oral corticosteroids

Osteoporosis agents (incl. bisphosphonates)

Investigator review of codes based on: https://www.cms.gov/icd10m/version37-fullcodecms/fullcode\_cms/P0244.html

Investigator review of codes based on:

https://pmc.ncbi.nlm.nih.gov/articles/PMC10478599/

 $Investigator\ review\ of\ codes\ based\ on: https://nccd.cdc.gov/ckd/Methods.aspx? Qnum=Q637, and the codes based on the code based on the code based on$ https://www.cms.gov/icd10m/FY2024-nprmversion41.0-fullcode\_cms/P2401.html Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/38527324/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/37796527/, https://pubmed.ncbi.nlm.nih.gov/35851329/,

https://pmc.ncbi.nlm.nih.gov/articles/PMC3985913/,

https://pubmed.ncbi.nlm.nih.gov/38503905/, https://pubmed.ncbi.nlm.nih.gov/35513234/

Investigator review of codes: https://pubmed.ncbi.nlm.nih.gov/36222554/, https://pubmed.ncbi.nlm.nih.gov/30287807/, https://pubmed.ncbi.nlm.nih.gov/22262606/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/36798959/, https://pubmed.ncbi.nlm.nih.gov/28438588/, https://pubmed.ncbi.nlm.nih.gov/31095068/Investigator review of codes: https://pubmed.ncbi.nlm.nih.gov/34624355/

Investigator review of codes Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK518983/ Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK278938/Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK513225/ Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK542331/ Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK576405/ Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK551656/, https://pmc.ncbi.nlm.nih.gov/articles/PMC4882495/, https://www.ncbi.nlm.nih.gov/books/NBK557848/ Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK518983/ Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK278938/

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK513225/Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK542331/ Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK576405/ Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK551656/, https://pmc.ncbi.nlm.nih.gov/articles/PMC4882495/,

https://www.ncbi.nlm.nih.gov/books/NBK557848/ Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/ Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK507904/ Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/ Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/lnvestigator review of codes, https://www.drugs.com,

https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/ Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK556025/ https://pubchem.ncbi.nlm.nih.gov/compound/441207

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/ Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/

Investigator review of codes

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/ Investigator review of codes, https://www.drugs.com,

https://www.ncbi.nlm.nih.gov/books/NBK482322/ (using class I and class II as class 2 is

beta blockers and class 4 is calcium channel blockers) Investigator review of codes, https://www.drugs.com, https://www.heart.org/en/health-

topics/cholesterol/prevention-and-treatment-of-high-cholesterol-

hyperlipidemia/cholesterol-medications

Investigator review of codes. https://www.drugs.com. https://www.heart.org/en/healthtopics/cholesterol/prevention-and-treatment-of-high-cholesterol-

hyperlipidemia/cholesterol-medications

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK537062/Investigator review of codes, https://www.drugs.com, https://www.ahajournals.org/doi/full/10.1161/JAHA.120.017559

Investigator review of codes, https://www.copdfoundation.org/Learn-More/I-am-a-Personwith-COPD/Treatments-Medications.aspx, https://getasthmahelp.org/medicationslist.aspx

Investigator review of codes, https://www.drugs.com,

https://www.ncbi.nlm.nih.gov/books/NBK547742/

Investigator review of codes, https://www.drugs.com, https://www.aaaai.org/tools-for-the-

public/drug-guide/oral-corticosteroid-medications Investigator review of codes based on: https://www.drugs.com,

https://www.ncbi.nlm.nih.gov/books/NBK470248/

Opioids

Anti-depressants Antipsychotics

Anxiolytics/hypnotics, benzodiazepines

Medication for dementia Urinary tract infections antibiotics

Laxatives

Number of distinct medications, median (iqr), mean (sd)

Number of office visits median (iqr), mean (sd)

Number of endocrinologist visits, median (iqr), mean (sd)

Number of cardiologist visits, median (iqr), mean (sd)

Number of internal medicine/family medicine visits, median (iqr), mean (sd)

Number of electrocardiograms, median (iqr), mean (sd)

Number of echocardiograms, median (iqr), mean (sd) Pharmacy out-of-pocket cost, median (iqr), mean (sd) Unique brand medications Unique generic medications Ratio of unique brand to generic medications

Colonoscopy/ Sigmoidoscopy

Flu vaccine / Pneumococcal vaccine

Pap smear test

PSA test

Fecal occult blood test Bone mineral density tests

Mammograms

Telemedicine

Number of HbA1c tests, median (iqr), mean (sd) Number of lipid panels, median (iqr), mean (sd) Number of creatinine tests, median (igr), mean (sd) Number of natriuretic peptide tests, median (iqr), mean (sd)

Number of urine tests, median (iqr), mean (sd)

HbA1c Glucose Creatinine

Systolic blood pressure Heart rate

**BMI** eGFR LDL HDL

Total cholesterol Triglycerides

Combined comorbidity score

Investigator review of codes, https://www.drugs.com,

https://pubmed.ncbi.nlm.nih.gov/31643200/#: -: text=They%20can%20also%20be%20information and the state of t

rmally,%2C%20codeine%2C%20oxycodone%2C%20hydrocodone%2C Investigator review of codes, https://www.drugs.com,

https://www.ncbi.nlm.nih.gov/books/NBK538182/

Investigator review of codes, https://www.drugs.com

Investigator review of codes, https://www.drugs.com, https://www.dea.gov/sites/default/files/2020-06/Benzodiazepenes-2020.pdf

https://www.ncbi.nlm.nih.gov/books/NBK470159/, https://www.drugs.com Investigator review of codes based on: https://www.drugs.com,

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7462122/,

https://go.drugbank.com/drugs/DB00382 https://pubmed.ncbi.nlm.nih.gov/35790044/

Investigator review of codes, https://www.drugs.com

N/A

https://www.cms.gov/files/document/mm13473-how-use-office-and-outpatient-

evaluation-and-management-visit-complexity-add-code-g2211.pdf,

https://www.cms.gov/files/document/physician-fee-schedule-pfs-payment-

officeoutpatient-evaluation-and-management-em-visits-fact-sheet.pdf
Data dictionary of Optum, Marketscan and https://www.cms.gov/Medicare/ProviderEnrollment-and-Certification/MedicareProviderSupEnroll/downloads/taxonomy.pdf,

https://www.cms.gov/medicare/provider-enrollment-and-

certification/medicareprovidersupenroll/downloads/taxonomycrosswalk.pdf Data dictionary of Optum, Marketscan and https://www.cms.gov/Medicare/Provider-

Enrollment-and-Certification/MedicareProviderSupEnroll/downloads/taxonomy.pdf,

https://www.cms.gov/medicare/provider-enrollment-and-

certification/medicareprovidersupenroll/downloads/taxonomycrosswalk.pdf Data dictionary of Optum, Marketscan and https://www.cms.gov/Medicare/Provider-

Enrollment-and-Certification/MedicareProviderSupEnroll/downloads/taxonomy.pdf,

https://www.cms.gov/medicare/provider-enrollment-and-

certification/medicareprovidersupenroll/downloads/taxonomycrosswalk.pdf

https://www.cms.gov/medicare-coverage-database/view/article.aspx?articleld=57326, https://firstcoastbillinggroup.com/ekg-billing-and-reimbursement/,

https://www.aapc.com/codes/coding-newsletters/my-cardiology-coding-alert/cpt-answer-5-common-ecg-coding-questions-175952-article

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8511132/,

https://pubmed.ncbi.nlm.nih.gov/34778785/, https://www.cms.gov/medicare-coverage-

database/view/article.aspx?articleid=56625&ver=27&,

https://www.medicalbillgurus.com/echocardiogram-cpt-code/

N/A

Investigator review of codes, https://www.drugs.com

Investigator review of codes, https://www.drugs.com Investigator review of codes, https://www.drugs.com

packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002

 $https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=refs%2Fheads%2Fcder_sir_wp002, https://www.cms.gov/medicare-coverage-database/view/article.aspx?articleld=54767&DocID=A54767, https://www.cms.gov/medicare-coverage-database/view/article.aspx.gov/medicare-coverage-database/vi$ 

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002, https://www.cms.gov/medicare-

coverage-database/view/article.aspx?articleId=54767&DocID=A54767

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002, http://www.icd9data.com/2012/Volume1/V01-V91/V70-V82/V72/default.htm,

http://www.icd9data.com/2012/Volume1/V01-V91/V70-V82/V76/default.htm

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-

packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002

Investigator review of codes

N/A

Investigator review of codes based on:

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002, https://www.cms.gov/medicare-

coverage-database/view/article.aspx?articleid=56448&ver=16&bc=0,

http://www.icd9data.com/2012/Volume1/V01-V91/V70-V82/V76/default.htm

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/33151319/,

https://www.cms.gov/newsroom/fact-sheets/medicare-telemedicine-health-care-provider-factsheet, https://www.aafp.org/family-physician/practice-and-career/getting-paid/coding/coding-

telehealth-audio-virtual-digital-visits.html https://pubmed.ncbi.nlm.nih.gov/34953068/

https://pubmed.ncbi.nlm.nih.gov/34953068/

https://pubmed.ncbi.nlm.nih.gov/34953068/

Investigator review of codes Investigator review of codes

N/A

N/A

N/A

N/A

N/A

N/A

N/A

N/A

N/A

A combined comorbidity score predicted mortality in elderly patients better than existing

scores, https://pubmed.ncbi.nlm.nih.gov/21208778/